BOS161721-02: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 In Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

ClinicalTrials.gov Identifier: NCT03371251

Final Protocol, Version 7.0 (Amendment 6), dated 30-April-2020 Final Protocol, Version 6.0 (Amendment 5), dated 23-July-2019 Final Protocol, Version 5.0 (Amendment 4), dated 23-January-2019 Final Protocol, Version 4.0 (Amendment 3), dated 27-July-2018 Final Protocol, Version 3.0 (Amendment 2), dated 21-March-2018 Final Protocol, Version 2.0 (Amendment 1), dated 08-November-2017 Final Protocol, Version 1.0, dated 06-October-2017

Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 30 April 2020; V7.0



# A RANDOMIZED DOUBLE-BLIND PHASE 1B/2 COMBINED STAGGERED MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF LIMITED STANDARD OF CARE

**SPONSOR** Boston Pharmaceuticals, Inc.

55 Cambridge Parkway, Suite 400

Cambridge, MA 02142

United States of America (USA)

INVESTIGATIONAL COMPOUND: BOS161721

PROTOCOL NUMBER: BOS161721-02

PHASE Phase 1b/2

INVESTIGATIONAL NEW DRUG (IND)

**NUMBER:** 

131796

ORIGINAL PROTOCOL DATE: 06 October 2017

**VERSION NUMBER:** V7.0 (Amendment 6)

VERSION DATE: 30 April 2020


## CLINICAL PROTOCOL APPROVAL FORM

| Protocol Title: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care. | |
|---|---|
| Study Number: BOS161721-02 | |
| Version | Date |
| Original Protocol | 06 October 2017 |
| Protocol Version 2.0 (Amendment 1) | 14 November 2017 |
| Protocol Version 3.0 (Amendment 2) | 21 March 2018 |
| Protocol Version 4.0 (Amendment 3) | 27 July 2018 |
| Protocol Version 5.0 (Amendment 4) | 23 January 2019 |
| Protocol Version 6.0 (Amendment 5) | 23 July 2019 |
| Protocol Version 7.0 (Amendment 6) | 30 April 2020 |

This study protocol was subject to critical review and has been approved by the sponsor. The information contained in this protocol is consistent with:

- The current risk-benefit evaluation of the investigational product
- The moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (Appendix 2), and principles of Good Clinical Practices (GCP) as described in 21 Code of Federal Regulations (CFR) parts 50, 54, 56 and 312 and according to applicable local requirements

The Investigator will be supplied with details of any significant or new findings, including adverse events, relating to treatment with the investigational product.

I agree with these statements and indicate my approval by signature for this protocol:

| Name and Title | Signature and Date |
|------------------------|--------------------|
| PPD , MD, PhD | PPD DocuSigned by: |
| Chief Medical Officer | |
| Boston Pharmaceuticals | |
| PPD , MD | DocuSigned by: |
| Vice President | PPD |
| Clinical Development | |
| Boston Pharmaceuticals | |




BOS161721-02

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care.


## CONFIDENTIALITY AND INVESTIGATOR STATEMENT

The information contained in this protocol and all other information relevant to BOS161721 are the confidential and proprietary information of Boston Pharmaceuticals, Inc., and except as may be required by federal, state, or local laws or regulation, may not be disclosed to others without prior written permission of Boston Pharmaceuticals, Inc.

I have read the protocol (Version 7.0, dated 30 April 2020), including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described. I will conduct this study as outlined herein, in accordance with the regulations stated in the Federal Code of Regulations for Good Clinical Practices and International Council for Harmonisation (ICH) guidelines, and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and any amendments, and access to all information provided by Boston Pharmaceuticals, Inc., or specified designees. I will discuss the material with them to ensure that they are fully informed about BOS161721 and the study.

| Principal Investiga | ator Name (printed) | Signature |
|---------------------|---------------------|-----------|
| Date | Site Number | |


# **PROTOCOL SUMMARY**

| Title: | A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care. |
|---|---|
| Indication | Adults with moderately to severely active SLE |
| Background and Rationale | Adults with moderately to severely active SLE SLE is a chronic systemic autoimmune disease with considerable heterogeneity in clinical manifestations and disease course. There is evidence that B- and T-cells are critical to the development of the disease, and that T-cell-derived cytokines such as interleukin-21 (IL-21) are involved in the SLE-associated inflammatory pathological response. BOS161721 is a humanized immunoglobulin G1 (IgG1) triple mutation monoclonal antibody (mAb) intended to have an extended terminal elimination half-life (t½) that selectively binds to and neutralizes IL-21, which acts on multiple cell types that drive inflammation and autoimmunity. In vivo, BOS161721 inhibits T-cell dependent antigen responses of B-cells and is being developed as a potential treatment for adults with moderately to severely active SLE. Nonclinical studies have evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), pharmacokinetics (PK), and immunogenicity of BOS161721 administered intravenously (IV) and subcutaneously (SC). The no observed adverse effect level (NOAEL) in Cynomolgus monkeys was determined to be 100 mg/kg (SC and IV), the highest dose tested. There were no injection site reactions in animals dosed subcutaneously. In a phase 1 single ascending dose (SAD) study, BOS161721 was administered IV and SC to healthy male and female adult subjects. This double-blind, placebo-controlled study evaluated 8 ascending dose levels (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) for safety, tolerability, PK, PD and immunogenicity. Overall, there were no clinically significant safety or tolerability findings from this study. Results from the phase 1 SAD study informed the dose regimens used for the multiple ascending doses (MAD) phase 1b portion of this trial. The MAD portion will involve 3 cohorts. The phase 2 portion will be a proof of concept (POC) part, where dose selection will be based on the data monitoring committee (DMC) and sponsor's assessment of safety, to |


Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 30 April 2020; V7.0

| Objectives | MAD Phase 1b | |
|---|---|---|
| and | OBJECTIVES | ENDPOINTS |
| Endpoints: | Primary | |
| | To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of adverse events (AEs) and serious adverse events (SAEs related AEs, AEs leading to study drug discontinuation, AE by severity and relatedness</li> <li>Injection site reactions</li> <li>Columbia Suicide Severity Rating Scale (C-SSRS)</li> <li>12-lead electrocardiograms (ECGs) parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> <li>Clinical laboratory results and change from baseline</li> <li>Physical examinations change from baseline</li> <li>Anti-drug antibodies (ADAs)</li> <li>Study drug exposure/compliance</li> </ul> |


# Secondary

 To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PD effects in patients with moderately to severely active SLE Pharmacokinetic Endpoints

- BOS161721 concentration by visit and time point
- Maximum observed concentration (C<sub>max</sub>), first time to maximum concentration (T<sub>max</sub>), area under the concentration-time curve (AUC), t½, systematic clearance (CL), volume of distribution (V<sub>d</sub>)

Pharmacodynamic Endpoints

- Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype
- Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit
- Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit







# POC Phase 2

| OBJECTIVES | ENDPOINTS |
|---|---|
| Prin | nary |
| To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on the SLE Responder Index 4 (SRI-4) | Primary Efficacy Endpoint The proportion of patients with a SRI-4 response at Day 210 (see Section 6.3.4.1) |


# Secondary

 To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment Secondary Efficacy Endpoints

- The proportion of patients with:
  - SRI-4 response at each visit
  - SRI-5 and SRI-6 response at each visit (Section 6.3.4.2)
  - a sustained reduction from baseline of oral corticosteroid (CS) (≤ 7.5 mg/day and < Day 0 dose) between Day 150 and Day 210
  - new or recurrent BILAG flares (≥ 1 qualifying BILAG A or > 1 qualifying BILAG B) through Day 210
  - PGA worsening
  - a BICLA response
  - a CLASI response
  - medication failures
- Changes and percent changes from baseline in:
  - CLASI
  - PGA
  - Total number of swollen joints, tender joints, and active joints (swelling and tenderness in the same joint) in the ACR-28 joint count
  - SLEDAI-2K
  - SLICC/ACR damage index
- Time to medication failure
- Group mean percent reduction in corticosteroid administration from baseline Day 0 dose through Day 210 in patients receiving ≥ 7.5 mg/day prednisone equivalent at Day 0
- Duration of longest SRI-4 response


Time to first BILAG flare (≥ 1 new or recurrent BILAG A or > 1 new or recurrent BILAG B) relative to baseline through Day 210 Safety To assess safety and Safety Endpoints tolerability of repeat Incidence and severity of doses of BOS161721 at adverse events (AEs) and the chosen dose serious adverse events administered SC in adult (SAEs), related AEs, AEs patients with moderately leading to study drug to severely active SLE on discontinuation, AEs by limited background severity and relatedness standard of care Injection site reactions treatment C-SSRS 12-lead ECGs parameter results at each visit and change from baseline Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline Clinical laboratory results and change from baseline Physical examinations changes from baseline ADAs Study drug exposure/compliance **Exploratory** 


270.




The MAD phase 1b portion of the study design will consist of 3 cohorts, with Cohort 1 containing 6 patients, where 5 of these patients will receive BOS161721 (active), and 1 will receive placebo. Cohorts 2 and 3 will each contain 12 patients, including 9 active and 3 placebo patients. Dose selection for each cohort is based on 90 day safety, tolerability, PK, and PD data review from the phase 1 SAD study (BOS161721-01) in healthy subjects. Each of the 3 doses (20, 60, and 120 mg) selected for the MAD portion are projected not to exceed the mean exposure of that achieved in the SAD study following the single 240 mg SC dose. Each patient may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

The MAD portion design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after the DMC evaluates the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after the DMC evaluation of the safety and tolerability data from Cohort 2 and Cohort 1. Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. This dose will not exceed doses tested during the MAD portion. For the POC portion, approximately 110 additional patients will be randomized to active or placebo groups in a 2:1 ratio. As in the MAD portion, each patient in the POC portion may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180. A maximum stable (for at least 6 weeks prior to Day 0) daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study. One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 120. Tapering of steroids during the course of the study will be highly encouraged and should be evaluated during the protocol-allowed tapering windows (Day 0 through Day 150) with the target of achieving a CS daily dose of ≤ 7.5 mg and < Day 0 dose between Day 150 and Day 210. Between Day 150 and Day 210, oral CS doses must be held constant due to the Day 210 endpoint evaluations. DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.

# Main Criteria for Inclusion and Exclusion

Inclusion Criteria:

1. Men and women, ages 18 to 70 years, inclusive


- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion OR Lupus nephritis as the sole clinical criterion in the presence of antinuclear antibodies [ANA] or anti-double-stranded deoxyribonucleic acid [dsDNA] antibodies), either sequentially or simultaneously
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA ≥ 1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
- 5. At screening, the total SLEDAI-2K score must be ≥ 8, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

- 6. A clinical SLEDAI-2K score of ≥ 6 at screening at Day 0. Clinical SLEDAI-2K score is defined as follows:
  - a. Contains points from arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, or vasculitis
  - Excludes parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive antidsDNA, decreased complement, thrombocytopenia, and leukopenia

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

- 7. Patients must have at least 1 qualifying A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system. If a BILAG B score is due to BILAG number 6, mild skin eruption, the CLASI activity score including erythema and scale/hypertrophy must be ≥ 3 excluding points from mucosal ulcers and alopecia
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 4.4


Note: Hips, shoulders, back, neck, and temporomandibular joints do not count towards the total number of joints with active synovitis. If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in at least 1 other body system for a total of 2 "B" BILAG body system scores.

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to Day 0) of the following permitted steroid-sparing agents:
    - Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. If AZA, myocophenolate mofetil, mycophenolic acid, hydroxychloroquine, or MTX were discontinued prior to screening, the washout period must be ≥ 12 weeks
  - Corticosteroids (prednisone or prednisone-equivalent) at a stable dose of up to 30 mg/day for at least 6 weeks prior to Day 0 (see Appendix 3)
    - For patients whose only SLE treatment is CSs, the stable CS dose must be ≥ 10 mg/day for at least 6 weeks prior to Day 0 and no more than 30 mg/day at the time of randomization
    - ii. Topical steroids may be used, but the dose must be stable for at least 6 weeks prior to Day 0. PRN topical steroids are not permitted
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening.
    Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding
  - Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

**Exclusion Criteria:** 

Patients presenting with any of the following will not be included in this study:

1. Drug-induced SLE, rather than "idiopathic" SLE


- 2. Other systemic autoimmune disease (e.g., erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic sclerosis, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON®-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed.
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS.
- 7. Concomitant illness that, in the opinion of the Investigator or the sponsor or their designee, is likely to require additional systemic glucocorticosteroid therapy during the study, (e.g., asthma), is exclusionary.
  - a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study.
- Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization.
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years.


- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
- 12. Cryptosporidium in the stool sample at screening.
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening.
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening.
- 15. CD4+ count < 150/µL at screening.
- 16. Platelets <  $50,000/\text{mm}^3$  ( $50 \times 10^9/\text{L}$ ) or <  $35,000/\text{mm}^3$  ( $35 \times 10^9/\text{L}$ ) if related to SLE, at screening.
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if related to SLE.
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol).
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 mL/minute based on Cockcroft-Gault calculation.
- 20. Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) > 2 × the upper limit of normal (ULN) at screening, unless explicitly related to lupus based on the Investigator's judgment.
- 21. Creatinine kinase (CK) > 3.0 × ULN at screening unless related to lupus myositis.
- 22. Total bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome).
- 23. Any other laboratory test results that, in the opinion of the Investigator or the sponsor or sponsor's designee, might place a patient at unacceptable risk for participating in this study.
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic mAb (e.g., IgG protein) or molecules made of components of mAbs.
- 25. History substance and/or alcohol abuse, or dependence within the past 1 year, at the Investigator's judgment.
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision).
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (e.g., cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, sponsor or sponsor's designee, would make the patient inappropriate for entry into this study.


- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial.
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer.
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 on the C-SSRS.
- 31. Current or pending incarceration.
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
- 33. Currently taking a total daily dose of > 30 mg morphine or morphine equivalent (see Appendix 7).
- 34. Body mass index (BMI)  $\geq$  40.0.

# Statistical Considerations

Below is a summary of the statistical methods. Further details can be found in Section 8.

Two analyses are planned: 1) an interim analysis to select the POC dose based on the MAD data; and 2) a final analysis at study completion. Additionally, DMC safety analyses will be performed for each MAD cohort and throughout the POC to monitor patient safety as described in the DMC charter. An additional analysis may be performed for the MAD portion of the study when all MAD patients have completed the safety follow-up, or withdrawn from the study, and prior to the final analysis. Data from the POC part of the study will be excluded from this additional analysis.

Unless stated otherwise, statistical testing will only be performed on the POC data and will be done using 2-sided overall alpha of 0.10. Data will be summarized descriptively by treatment and overall for each study phase. For the MAD portion, BOS161721 will be summarized overall and by each dose level and placebo patients from each cohort will be combined.

The descriptive summaries for the categorical data will include number and percentage. The descriptive summaries for the continuous data will include number, mean, median, standard deviations (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, median, and maximum. Counts, medians, 25<sup>th</sup> and 75<sup>th</sup> percentiles, and standard error will be presented for time-to-event data.


All safety analyses will be performed using the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. All efficacy analyses will be performed using the full analysis set (FAS), defined as all patients who receive at least 1 dose of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. Select efficacy analyses may also be performed on the per protocol (PP) set.

Binary efficacy endpoints, including the primary efficacy endpoint, will be assessed via Pearson's chi-squared analysis.

Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) when applicable, adjusting for the baseline value. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test.

Adverse event data will be coded to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be summarized, based on coded terms, using frequency and percentage of patients. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters, will be summarized at each individual visit.


# **TABLE OF CONTENTS**

| A RANDOMIZED DOUBLE-BLIND PHASE 1B/2 COMBINED STAGGERED MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF LIMITED STANDARD OF CARE | 4 |
|---|---|
| CLINICAL PROTOCOL APPROVAL FORM | |
| CONFIDENTIALITY AND INVESTIGATOR STATEMENT | |
| PROTOCOL SUMMARY | |
| TABLE OF CONTENTS | |
| LIST OF IN-TEXT TABLES | |
| LIST OF IN-TEXT FIGURES | |
| LIST OF ABBREVIATIONS | |
| 1 INTRODUCTION AND RATIONALE | |
| 1.1 Indication | 29 |
| 1.2 Background and Rationale | 29 |
| 1.2.1 Overview of the Disease State | <b>2</b> 9 |
| 1.2.2 BOS161721 Development | <mark>2</mark> 9 |
| 1.2.2.1 Interleukin-21 | 30 |
| 1.2.2.2 Preclinical Studies | 31 |
| 1.2.2.3 Clinical Studies | 33 |
| 1.2.3 Study Dose Selection | 33 |
| 1.2.4 Risk-Benefit Assessment | 35 |
| 1.2.5 Potential Risks | 35 |
| 1.2.5.1 Anaphylaxis and Serious Allergic Reactions | |
| 1.2.5.2 Injection Site Reactions | |
| 1.2.5.3 Immune Complex Disease | |
| 1.2.5.4 Infections | |
| 1.2.5.5 Malignancy | |
| 1.2.5.6 Hepatic Function Abnormality | |
| 1.2.5.7 Failure of Vaccination | |
| 1.2.5.8 Potential for Drug-Drug Interactions | |
| 1.2.5.9 Potential Risk to Fetal Development | |
| 2 STUDY OBJECTIVES AND ENDPOINTS | |
| 2.1 Phase 1b Multiple Ascending Dose | |
| 2.2 Phase 2 Proof of Concept | |
| 3 STUDY PLAN | |
| 3.1 Study Design | |
| 3.1.1 Multiple Ascending Dose Phase 1b | |
| 3.1.1.1 Dose Escalation for the MAD Portion | |
| 3.1.1.2 Dose Limiting Toxicity (DLT) | 44 |

Protocol Date and Version: 30 April 2020; V7. 0

| | 540 B | |
|---|---|---|
| 3.1.1.3 | | |
| 3.1.2 | POC Phase 2 | |
| 3.1.2.1 | BOS161721 POC Dose Selection and Justification | |
| 3.1.2.2 | , | |
| | Randomization and Blinding | |
| | Study Schematic | |
| | Schedule of Assessments | |
| | End of Study | |
| | PULATION | |
| | Participant Recruitment | |
| | Number of Patients | |
| | Patient Screening | |
| | Inclusion Criteria | |
| | Exclusion Criteria | |
| | Concomitant Medications | |
| 4.6.1 | Corticosteroid | |
| 4.6.2 | Other Prohibited and/or Restricted Treatments | |
| | Women of Childbearing Potential | |
| 4.7.1 | Determination of Menopause | |
| 4.7.2 | Contraception | |
| | Deviation from Inclusion/Exclusion Criteria | |
| 4.8.1 | Patient Withdrawal and Replacement | |
| | UDY PROCEDURES | |
| | Screening | |
| 5.1.1 | Retesting During Screening Period | |
| | Enrollment/Randomization and Day 0 Treatment | |
| | Treatment Period/Follow-Up Visits | |
| | Safety Follow-Up VisitsPremature Discontinuation | |
| | Contingency Plans During the COVID-19 Pandemic | |
| | SESSMENTS Medical History, Demographic and Other Baseline Information | |
| 6.2.1 | Safety Assessments | |
| 6.2.1.1 | • | |
| 6.2.1.1 | Pregnancy testing | |
| 6.2.2 | • | |
| 6.2.2.1 | Adverse Events | |
| 6.2.2.1 | Definitions Recording of Adverse Events | |
| 6.2.2.3 | <del>_</del> | |
| 6.2.2.4 | | |
| 0.4.4.4 | Causality of Auverse Everits | 13 |

| Cli | nica | l Study | Protoco | l: B | OS1617 | 721-02 | |
|-----|------|---------|---------|------|--------|--------|----|
| _ | | | | | | | ٠. |


| | · | |
|--------|--------------------------------------------------------------|----|
| 6.2.2. | 5 Seriousness of Adverse Events | 74 |
| 6.2.2. | 6 Adverse Events of Special Interest | 74 |
| 6.2.2. | 7 Reporting of Adverse Events | 77 |
| 6.2.2. | 8 Follow Up of Adverse Events | 79 |
| 6.2.3 | Vital Signs | 80 |
| 6.2.4 | 12-Lead Electrocardiograms | 80 |
| 6.2.5 | Physical Examinations | |
| 6.2.6 | C-SSRS | 80 |
| 6.2.7 | Injection Site Reactions | 81 |
| 6.2.8 | Immunogenicity | 81 |
| 6.3 | Efficacy Assessments | 81 |
| 6.3.1 | SLEDAI-2K | 81 |
| 6.3.2 | BILAG 2004 | 82 |
| 6.3.3 | PGA of Disease Activity | 82 |
| 6.3.4 | Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response | 82 |
| 6.3.4. | | |
| 6.3.4. | 2 SRI-5 and SRI-6 Response | 83 |
| 6.3.4. | 3 BICLA Response | 83 |
| 6.3.5 | CLASI Response | 83 |
| 6.3.6 | ACR-28 Joint Count | 83 |
| 6.4 | Other Variables | 83 |
| 6.4.1 | SLICC/ACR Damage Index | 83 |
| 6.4.2 | PROs | 84 |
| 6.5 | Pharmacokinetic Assessments | 84 |
| 6.6 | Pharmacodynamic Assessments | 84 |
| 6.7 | Pharmacokinetic/Pharmacodynamic Relationship | 84 |
| 6.8 | Protocol Deviations | 85 |
| 7 S | TUDY DRUG MANAGEMENT | 85 |
| 7.1 | Description | 85 |
| 7.1.1 | Formulation | 85 |
| 7.1.2 | Storage | 85 |
| 7.2 | Packaging and Shipment | 85 |
| 7.3 | Dose and Administration | 85 |
| 7.4 | Accountability | 86 |
| 7.5 | Prohibited Concomitant Therapy | 86 |
| 7.6 | Compliance | 86 |
| 8 S | TATISTICS | 86 |
| 8.1 | Sample Size | 87 |
| 8.2 | Statistical Methods | 88 |
| 8.2.1 | Analysis Populations | |
| 8.2.2 | Demographics and Baseline Characteristics | 88 |

| Clinical Study Protocol: BOS161721-02 |
|-------------------------------------------------|
| Protocol Date and Version: 30 April 2020: V7. 0 |

| 1 101000 | of Bate and Version. 66 April 2026, V1. 6 | |
|---|---|---|
| 8.2.3 | Primary Efficacy Endpoint(s) | 89 |
| 8.2.4 | Secondary Efficacy Endpoint(s) | 89 |
| 8.2.5 | Analysis of Safety | |
| 8.2.5. | 1 Safety Analysis | 89 |
| 8.2.6 | Pharmacokinetic and Pharmacodynamic Data | 90 |
| 8.2.6. | 1 Analysis of Pharmacokinetic Data | 90 |
| 8.2.6.2 | 2 Analysis of Pharmacodynamic Data | 90 |
| 8.2.6.3 | Population Pharmacokinetic Analysis or PK/PD Modeling | 90 |
| 8.3 | Interim Analysis and Power | 90 |
| 9 E | THICS AND RESPONSIBILITIES | 91 |
| 9.1 | Good Clinical Practice | 91 |
| 9.2 | DMC | 91 |
| 9.3 | Institutional Review Board/Independent Ethics Committee | 92 |
| 9.4 | Informed Consent | 92 |
| 9.5 | Records Management | 92 |
| 9.6 | Source Documentation | 93 |
| 9.7 | Study Files and Record Retention | 93 |
| 10 Al | UDITING AND MONITORING | 94 |
| 11 A | MENDMENTS | 94 |
| 12 S | TUDY REPORT AND PUBLICATIONS | 95 |
| 13 S | TUDY DISCONTINUATION | 95 |
| 14 C | ONFIDENTIALITY | 95 |
| 15 RI | EFERENCES | 96 |
| 16 AF | PPENDICES | . 100 |
| 16.1 | Appendix 1: Names of Study Personnel | . 101 |
| 16.2 | Appendix 2: Declaration of Helsinki | . 102 |
| 16.3 | Appendix 3: Commonly Used Corticosteroid Equivalents | . 107 |
| 16.4 | Appendix 4: Medication Washout Periods | . 108 |
| 16.5 | Appendix 5: BILAG-2004 (Study-Specific Modified Criteria) | . 109 |
| 16.6 | Appendix 6: Injection Site Reaction Grading Scale | . 110 |
| 16.7 | Appendix 7: Opioid Oral Morphine mg Equivalents of Commonly Used | |
| | Opioids | . 111 |
| 16.8 | Appendix 8: Schedule of Assessments - Phase 1b Multiple Ascending Dose | 114 |
| 16.9 | Appendix 9: Protocol Summary of Changes | |
| | LIST OF IN-TEXT TABLES | |
| Table | Schedule of Assessments - Phase 2 Proof of Concept (POC) | 49 |
| Table | | |
| Table | 3. Causality Definitions | 73 |


| | Boston Pharmaceuticals, Ind<br>v Protocol: BOS161721-02<br>e and Version: 30 April 2020; V7. 0 |
|---|---|
| Table 4. | Schedule of Assessments - Phase 1b - Multiple Ascending Dose 114 |
| LIST OF IN-TEXT FIGURES | |
| Figure 1. | Individual pSTAT3 C <sub>min</sub> Levels Versus Dose |

Figure 2.


Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 30 April 2020; V7. 0

### LIST OF ABBREVIATIONS

ACR American College of Rheumatology

ADA anti-drug antibody
ADL activities of daily living

AE adverse event

AIDS acquired immune deficiency syndrome

ALT alanine aminotransferase
ANA antinuclear antibodies
ANC absolute neutrophil count

ANOVA analysis of variance
ANCOVA analysis of covariance

APL antiphospholipid

AST aspartate aminotransferase

AUC area under the concentration-time curve

AZA azathioprine

BICLA BILAG-based Composite Lupus Assessment

BILAG British Isles Lupus Assessment Group

BMI body mass index BP blood pressure

BUN blood urea nitrogen

BW body weight C complement

C-SSRS Columbia Suicide Severity Rating Scale

CD cluster of differentiation

CK creatine kinase

CL systematic clearance

CLASI Cutaneous Lupus Erythematosus Area and Severity Index

C<sub>max</sub> maximum plasma concentration

CMH Cochran-Mantel-Haenszel

CS corticosteroids

CSR clinical study report

DILI drug-induced liver injury

DLT dose-limiting toxicity

DMC data monitoring committee

dsDNA double-stranded deoxyribonucleic acid


ECG electrocardiogram
EOT end of treatment

eCRF electronic case report form

F female

CCI

FAS full analysis set

Fc fragment crystallizable

FDA Food and Drug Administration FSH follicle stimulating hormone

GCP Good Clinical Practice

eGFR estimated glomerular filtration rate

GLP Good Laboratory Practice

GWAS genome-wide association studies

γc gamma chain HBV hepatitis B virus

hCG human chorionic gonadotropin

HCI hydrochloride HCV hepatitis C virus

HIV human immunodeficiency virus

HR heart rate

HRT hormone replacement therapy

IA interim analysis

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonization

IEC Independent Ethics Committee

lg immunoglobulin

IL interleukin

IL-21R interleukin 21 receptor

IM intramuscular

IFNy interferon gamma

INR International Normalized Ratio
IRB Institutional Review Board

IUD intrauterine device

IV intravenous

IWRS interactive web response system


JAK Janus kinase

kg kilogram

KLH keyhole limpet hemocyanin LOCF last observation carried forward

M male

mAb monoclonal antibody
MAD multiple ascending dose

MAPK mitogen-activated protein kinase

MedDRA Medical Dictionary of Regulatory Activities

MS multiple sclerosis
MTX methotrexate

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse

**Events** 

NIAID/FAAN National Institute of Allergy and Infectious Diseases/Food Allergy and

Anaphylaxis Network

NK natural killer

NOAEL no observed adverse event level

NO nitric oxide

NSAID nonsteroidal anti-inflammatory drug

OTC over-the-counter
PD pharmacodynamics
PEF peak expiratory flow

PGA Physician's Global Assessment

PK pharmacokinetics
POC proof of concept
PP per protocol

PR (interval) from onset of the p-wave to the end of the r-wave

pSS primary Sjögren's syndrome

pSTAT3 phosphorylated signal transducer and activator of transcription 3

PT preferred term

QRS (interval) from the onset of the q-wave to the end of the s-wave QT (interval) from onset of the QRS complex to the end of the T wave

QTcF QT interval corrected for heart rate using Fridericia's formula

QFT-G QuantiFERON®-TB Gold In-Tube

RA rheumatoid arthritis


RR (interval) from the onset of the r-wave to the onset of the next

consecutive r-wave

SAD single ascending dose
SAE serious adverse event
SAP statistical analysis plan

SC subcutaneous

SDMT safety data monitoring board

CCI

SLE systemic lupus erythematosus SLEDAI-2K SLE Disease Activity Index 2000

SLICC Systemic Lupus International Collaborating Clinics

Sm Smith

SOC system organ class

SRI-4 SLE Responder Index 4
SRI-5 SLE Responder Index 5
SRI-6 SLE Responder Index 6

SS safety analysis set

SSA Sjögren syndrome-A (Ro) SSB Sjögren syndrome-B (La)

STAT3 signal transducer and activator of transcription 3 SUSAR suspected unexpected serious adverse reaction

ty<sub>2</sub> terminal elimination half-life

TB tuberculosis

TDAR T-cell dependent antibody response

Tfh T-follicular helper

Th T-helper

TK toxicokinetics

T<sub>max</sub> first time to maximum concentration

Treg regulatory T-cell

ULN upper limit of normal

US United States

V<sub>d</sub> volume of distribution

WBC white blood cell

WHO World Health Organization

WOCBP women of childbearing potential

YTE triple mutation


# 1 INTRODUCTION AND RATIONALE

#### 1.1 Indication

BOS161721 is a humanized monoclonal antibody (mAb), which binds to and inhibits interleukin-21 (IL-21) bioactivity, and is being developed for the treatment of moderately to severely active systemic lupus erythematosus (SLE) in adults.

# 1.2 Background and Rationale

#### 1.2.1 Overview of the Disease State

SLE is a chronic inflammatory autoimmune disease that has variable manifestations in multiple organ systems and follows a relapsing and remitting course. The disease process includes abnormal immune responses mediated by tissue-binding autoantibodies and immune complex deposition, giving rise to tissue damage often resulting in end organ disease and even mortality. Survival of SLE has improved due to earlier detection, improved overall medical care, and standardized SLE treatment with corticosteroids (CS), immunosuppressants, and cytotoxic agents. However, some of the morbidity in patients with SLE is related to its treatment. Comparison of early and late outcomes in patients with SLE demonstrate that death in early disease is most commonly due to infections and active SLE causing multi-system organ damage, while thromboses were the most common cause of death during later disease.<sup>2</sup>

The reported prevalence of SLE in the United States (US) is 20 to 70 cases per 100,000 people.<sup>3</sup> More than 90% of cases of SLE occur in women, frequently starting at childbearing age. Women of color are disproportionately affected by SLE. This suggests multiple genetic and environmental factors are at play. Accordingly, a multifactorial view of the immunopathogenesis of SLE suggests more than 1 area of interest, including breach in central tolerance in the adaptive arm of the immune system, peripheral amplification of the autoimmune response by the innate immune system, and local processes in the target organ that facilitate end-organ disease.<sup>4</sup>

# 1.2.2 BOS161721 Development

Boston Pharmaceuticals is developing BOS161721 for the treatment of SLE. BOS161721 is a humanized immunoglobulin G1 (IgG1) mAb with extended half-life directed against human IL-21.

Murine mAb 19E3, the progenitor of BOS161721, was generated using mouse hybridoma technology.19E3 has subpicomolar (pM) affinity to human IL-21 and was selected for its potent neutralization of IL-21 bioactivity. BOS161721 was generated by the humanization of mAb 19E3 where its complementarity-determining regions were grafted onto a human IgG1 kappa backbone. The fragment crystallizable (Fc) portion of BOS161721 contains a YTE (M252Y/S254T/T256E triple mutation) in the constant domain of the IgG1 heavy chain that was introduced into the parental molecule, 19E3, intended to prolong the in vivo terminal elimination half-life (t½) of the mAb.<sup>5</sup> Thus,


Clinical Study Protocol: BOS161721-02


BOS161721 retains sub-pM binding to IL-21 and prevents IL-21 from binding to the IL-21 receptor (IL-21R), inhibiting IL-21 bioactivity.

BOS161721 binds to human IL-21 and Cynomolgus monkey IL-21, which are highly homologous, and neutralizes the bioactivity of both. BOS161721 is specific for IL-21 as it does not bind to or inhibit the other gamma-chain (γc) family of cytokines, and acts to specifically neutralize the IL-21 pathway. In in vitro studies, BOS161721 inhibited downstream IL-21-induced signaling, IL-21-induced plasma cell differentiation, and IL-21-induced natural killer (NK) cell activation. In in vivo studies, BOS161721 significantly inhibited the T-cell dependent antibody response (TDAR) to immunization with a protein antigen as well as B-cell expansion following a second protein antigen immunization in Cynomolgus monkeys.

#### 1.2.2.1 Interleukin-21

IL-21 is an inflammatory cytokine, which belongs to a family of cytokines that also includes IL-2, IL-4, IL-7, IL-9, and IL-15, all of which bind to private receptors in complex with the common cytokine receptor yc.6 Most cytokines in this family are critically important for both the maintenance and function of T-cell and B-cell responses. IL-21 signals through a receptor complex consisting of its own private receptor, the IL-21R and yc.<sup>6,7</sup> Engagement of the IL-21R/yc complex leads to the activation of several signaling pathways, including the Janus kinase/signal transducer and activator of transcription, mitogen-activated protein kinase (MAPK) and phosphoinositide 3-kinase pathways.8 IL-21 is produced mainly by T-cells and NK T-cells, but neutrophils have also been reported to produce IL-21.9,10 The IL-21R is expressed on a broad array of cell types, including B-cells, T-cells, NK-cells, macrophages and dendritic cells, as well as other hematopoietic and nonhematopoietic cells such as fibroblasts, keratinocytes, and intestinal epithelial cells. 9,11 Activation of signal transducer and activator of transcription 3 (STAT3) via phosphorylation is critical in regulating human B-cell responses to IL-21<sup>12</sup>; phosphorylated STAT3 (pSTAT3) forms a homodimer, which translocates to the nucleus where it initiates transcription of the IL-21 gene, forming an autocrine loop for IL-21 production via STAT3 phosphorylation. 13 In addition, IL-21 has been shown to upregulate expression of its own receptor<sup>14</sup> and induces an autocrine feedback loop. 15

IL-21 modulates various aspects of immune function. It promotes cluster of differentiation 4 (CD4+) T-cell differentiation and promotes the generation of T-helper (Th)17<sup>16</sup> and T-follicular helper (Tfh) cells.<sup>15,17</sup> In mice, IL-21 has been shown to regulate the balance between Th17 and regulatory T-cell (Treg), in that it increases Th17, while inhibiting Treg differentiation.<sup>18</sup> Less is understood with regards to human Tregs, although IL-21 has been reported to counteract Treg suppression of human effector T-cells<sup>19</sup> and blockade of IL-21 promotes Treg generation in a murine model of graft versus host disease induced by human T-cells.<sup>20</sup> IL-21 upregulates CD8+ T-cell and NK-cell expansion and cytolytic activity by increasing granzyme B and perforin.<sup>21,22</sup> IL-21 also has been reported to increase granzyme B in plasmacytoid dendritic cells and B-cells resulting in inhibition of T-cell responses.<sup>23,24</sup> IL-21 also has a variety of


Clinical Study Protocol: BOS161721-02


effects on nonhematopoietic cells, such as stromal cells and induces inflammation through matrix metalloproteinase release by gut intestinal fibroblasts.<sup>25</sup>

One principal non-redundant role of IL-21 is the promotion of B-cell activation, differentiation, or death during humoral immune responses.<sup>14</sup> Furthermore, increased IL-21 production is characteristic of several autoimmune diseases and is likely to contribute to autoantibody production as well as pathologic features of autoimmune disease.<sup>26</sup> The critical role of IL-21 in promoting humoral and other immune responses makes it an important focus of potential therapeutic interventions in conditions characterized by overproduction of pathogenic autoantibodies. IL-21 production by Tfh cells in humans is believed to play a major role in driving the autoantibody production through its role in plasma cell differentiation. Importantly, Tfh cell populations are expanded in patients with autoimmune diseases such as lupus, bullous pemphigoid, rheumatoid arthritis (RA) and primary Sjögren's syndrome (pSS) and have been reported to correlate with IL-21 levels, autoantibodies, and disease severity. 26,27,28,29 Furthermore, loss of number and functionality of Tregs has been associated with autoimmune diseases such as SLE and giant cell arteritis, which IL-21 is expected to modulate. 30,31 Thus, neutralization of IL-21 in settings of autoimmunity is expected to impact several cell populations believed to be involved in the pathogenesis of autoimmune disorders including SLE.

BOS161721 selectively binds IL-21 with high affinity to neutralize IL-21, and due to its pleiotropic nature, neutralization of IL-21 is expected to impact several cell populations believed to be involved in the pathogenesis of SLE. Importantly, patients with SLE have elevated IL-21 plasma levels that correlate with the severity of the disease. Recently, genome-wide association studies (GWAS) have provided convincing evidence that the chromosomal 4q 27 region harbors the IL-21 genes and is associated with chronic inflammatory disorders, including SLE.<sup>29</sup>

#### 1.2.2.2 Preclinical Studies

The pharmacokinetics (PK) of BOS161721 were characterized following single-dose intravenous (IV) administration of BOS161721 (0.01 to 30 mg/kg) in male Cynomolgus monkeys or repeat, every 2 weeks IV administration (15 to 100 mg/kg) and subcutaneous (SC) administration (50 mg/kg) in male and female Cynomolgus monkeys. Systemic exposure was approximately dose-proportional within the tested dose range. SC bioavailability was determined to be 64.3%.

Two single-dose (IV) non-good laboratory practice (GLP) studies conducted in Cynomolgus monkeys evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), and immunogenicity of BOS161721. Following a single IV administration (slow bolus), there were no BOS161721-related adverse changes, resulting in a no-observed-adverse-effect-level (NOAEL) value of 30 mg/kg, the highest dose tested among 2 studies.


| In a repeat-dose GLP toxicology study in Cynomolgus monkey | vs ROS161721 was |
|---|---|
| administered every 2 weeks by IV or SC (50 mg/kg) administration of 7 doses). | |
| 51 7 do3c3). <mark>col</mark> | |
| | The |
| NOAEL was determined to be 100 mg/kg (SC and IV), the high | . The nest dose tested. |
| An additional GLP, repeat-dose toxicity study was conducted in<br>(4 males and 4 females per dose group) following every 2 wee<br>by SC (10, 30, and 100 mg/kg) injection for a total of 14 doses | ks (Q2W) administration |
| | There were |
| no BOS161721-related effects on survival, clinical signs, male ophthalmologic parameters, electrocardiogram (ECG) findings macroscopic observations, organ weights, or microscopic obse | , clinical pathology, |
| the NOAEL CO | The 100 mg/kg/dose was |
| the NOAEL CCI | |


#### 1.2.2.3 Clinical Studies

BOS161721-01 was a double-blind, phase 1, single ascending dose (SAD) study to assess the safety, PK, and PD of BOS161721 in healthy subjects. The primary objective of the study was to characterize the safety and tolerability of IV and SC SADs of BOS161721 in an otherwise healthy subject population without concomitant illnesses, immune abnormalities, or concomitant medications. Secondary objectives included characterization of the PK and immunogenicity of BOS161721, and exploratory objectives included the evaluation of the effect of BOS161721 on TDAR to keyhole limpet hemocyanin (KLH) (primary and secondary immunizations) in healthy subjects, the effects of BOS161721 on plasma levels of IL-21 (free and bound), and the evaluation of the effect of BOS161721 on IL-21 gene expression (via gene signature) in blood. This study consisted of 8 cohorts. Subjects were randomized in a 3:1 ratio (BOS161721: placebo) and received either a single dose of BOS161721 (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) or placebo, with safety follow-up. For the first cohort, after the first 2 subjects were dosed (1 active and 1 placebo), there was a minimum gap of 48 hours before the remaining subjects from that cohort were dosed, to allow for an initial review of any emerging safety and tolerability data. For all cohorts, escalation to the next dose was not sooner than 8 days after all the subjects in the prior cohort had been dosed and were based on a review of at least 7 days of safety and tolerability data by the Safety Data Monitoring Team (SDMT).

Blood samples were collected at every in-house study visit for BOS161721 concentration determinations. Blood samples were also collected for determination of IL-21 plasma levels (free and total). Safety was assessed based on the occurrence of treatment-emergent AEs, hepatic function abnormality, and acute and delayed hypersensitivity reactions. Other safety variables included ECGs, vital signs (blood pressure [BP], heart rate, and temperature), safety laboratory assessments, blood sampling for ADAs, total IgG and immunoglobulin M (IgM) levels, CD4+ count, and full and targeted physical examinations. Overall, there were no clinically significant findings from this study. Adverse events reported as related to the study drug, particularly infections, were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. There was 1 serious adverse event (SAE; death due to pulmonary embolism) that occurred 127 days after a single administration of 240 mg SC dose of BOS161721. The causality of this single SAE was not attributed to study drug and further information can be found in the Investigator's Brochure. Final PK data from the SAD study demonstrates BOS161721 has a mean t1/2 ranging from 80 to 87 days for doses of ≥ 30 mg in healthy subjects.

# 1.2.3 Study Dose Selection

Doses have been selected for the multiple ascending dose (MAD) phase 1b portion based on a 90 day safety, tolerability, PK, and PD data review from the phase 1 SAD study (BOS161721-01); the SDMT reviewed the blinded safety data from subjects for each dose cohort (8 cohorts, evaluating 1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg), along with the accumulated safety and available PK/PD data


from all subjects in the previous dose cohorts, to make a decision on whether to proceed to the next higher dose level, repeat a dose level, or stop dose escalation. Overall, there were no clinically significant safety or tolerability findings from this study.

Based on the Day-90 interim cut of the PK and biomarker data in the BOS161721-01 study, the recommended doses for evaluation in the MAD portion of this study are 20, 60, and 120 mg SC monthly. This dose recommendation is supported by evidence of linear PK with BOS161721 resulting in a median first time to maximum concentration (T<sub>max</sub>) of 6 days and an apparent terminal half-life of 44 days. Furthermore, pSTAT3 suppression, a marker of IL-21 target engagement, follows a similar time course of the mAb levels, with maximal and sustained suppression apparent with doses greater than 30 mg SC (Figure 1).



Figure 1. Individual pSTAT3 Cmin Levels Versus Dose

IV = intravenous, pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SC = subcutaneous

All doses selected for the MAD portion are projected not to exceed the mean exposure of that achieved following the highest single dose of 240 mg SC administered in the phase 1 SAD study. Cohort 1 will include randomized treatment to the 20 mg dose. Based on the staggered study design, the data monitoring committee (DMC) will perform a scheduled review of safety data and sequentially consider dose escalation for Cohorts 2 and 3. In addition, the DMC and Boston Pharmaceuticals will conduct a data


Clinical Study Protocol: BOS161721-02


review to determine which dose will be carried forward into the proof of concept (POC) phase 2 portion. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD portion (see Section 3.1.2.1 for the chosen POC dose and justification).

#### 1.2.4 Risk-Benefit Assessment

The available preclinical data on BOS161721, the findings in clinical study BOS161721-01, and existing clinical information on IL-21 inhibitors suggest that the present clinical study has an acceptable risk-benefit ratio. In this study, the risk-benefit assessment of BOS161721 in adult patients with moderately to severely active SLE will be ongoing, with step-wise evaluations during the staggered MAD portion. The DMC used in this study is charged with assessing such actions in light of an acceptable benefit-risk profile for BOS161721 as an anti-IL-21 mAb. Formal DMC monitoring meetings will occur as described in the DMC Charter. Two weeks after Cohort 1 has received a second dose of study drug, the DMC will evaluate the safety and tolerability data from Cohort 1 to determine the recommended dose for Cohort 2. Two weeks after 8 patients in Cohort 2 receive a second dose, the DMC will determine if dose escalation to Cohort 3 can proceed. Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3 during the MAD part of study. Thereafter, DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter. With the agreement of the DMC and sponsor, this schedule may be modified depending on the rate of patient accrual. Additional details can be found in the DMC Charter.

The benefit of participation for all patients in this study is close monitoring of their medical condition and safety of their treatment. Those randomized to the active treatment arm may potentially experience improvement in their SLE disease. Those randomized to the placebo (in combination with standard of care) arm are not expected to obtain any additional benefit, beyond those of their background treatment, though close monitoring of their medical condition and safety may itself be associated with improving their SLE.

#### 1.2.5 Potential Risks

Potential risks based on the mechanism of action of BOS161721 include infections, risks associated with the administration of any foreign protein or biologic agent, including injection site reaction, anaphylaxis, serious allergic reaction, and development of ADAs. ADAs could result in immune complex disease (with manifestations such as arthralgias, serum-sickness, and vasculitis), or altered BOS161721 levels or activity. Further details can be found in the current Investigator's Brochure (IB) for BOS161721, which contains comprehensive toxicology, preclinical and clinical information on BOS161721.


Two investigational drug products are considered to be in the same pharmacological class as BOS161721 based on interruption of signaling through the IL-21 signaling pathway. No potential risk generalizable across the class has been observed with these investigational products. Based on the clinical phase 1 SAD study (BOS161721-01), AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc.), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs.

The majority of IgG elimination occurs via intracellular catabolism, following fluid-phase or receptor-mediated endocytosis. This type of endocytosis and elimination is a form of target-mediated disposition where the interaction of the drug and its pharmacological target (e.g., a target receptor) serves as a significant contributor to the kinetics of antibody distribution and elimination. Renal elimination, which is a primary pathway of clearance of small-molecule drugs, is relatively unimportant for IgG, as its large size prevents efficient filtration through the glomerulus. Secretion into the bile is an important pathway of elimination of IgA antibodies, but this route is not a significant contributor to the elimination of IgG antibodies. Thus, risk to renal and hepatic systems due to metabolism of BOS161721 is low.<sup>33</sup>

### 1.2.5.1 Anaphylaxis and Serious Allergic Reactions

As with the administration of any foreign protein and/or other biological agents, acute hypersensitivity reactions, including acute anaphylactic/hypersensitivity, severe allergic, and anaphylactoid reactions may follow infusion of mAbs and can be caused by various mechanisms. These acute hypersensitivity reactions may be severe and result in death.

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria,<sup>34</sup> and are discussed in Section 6.2.2.6.1.

Based on the phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed.

Patients with a known history of allergy or severe hypersensitivity reaction to any component of BOS161721 formulation or patients with a history of anaphylaxis to any other biological therapy such as mAbs will be excluded from studies with BOS161721. In addition, appropriate drugs and medical equipment to treat acute hypotensive, bronchoconstrictive, or anaphylactic reactions will be immediately available at the unit and study personnel will be trained to recognize and treat these reactions.

#### 1.2.5.2 Injection Site Reactions

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC for 3 months (a total of 7 doses). There were no injection site reactions in animals dosed subcutaneously. Further, there were no reports of injection site reactions in the 26-week GLP toxicology study in Cynomolgus monkeys.


Based on the phase 1 SAD study (BOS161721-01), incidence of injection site reactions in subjects who received BOS161721 was similar to placebo.

Patients will be monitored for local injection site reactions in this study (see Section 6.2.7).

### 1.2.5.3 Immune Complex Disease

The potential risk of immune complex disease for BOS161721 is theoretical, based on the known risks associated with mAbs. The administration of a mAb can result in the formation of ADAs. Administration of the mAb in the presence of ADA may result in the formation of circulating antibody-antigen complexes potentially resulting in altered BOS161721 levels or activity or deposition of the complexes in microvasculature. Complement is frequently involved in the latter setting, and the breakdown products of complement attract polymorphonuclear leukocytes to the site of deposition where they can provoke local tissue damage through specific or nonspecific release of enzymes. Two of the more common end-organ targets are the blood vessels (vasculitis) and kidney (nephritis). These clinical manifestations represent immune complex disease or Type III hypersensitivity. Although BOS161721 is a humanized mAb, ADAs may develop; however, the likelihood of occurrence of immune complex disease with BOS161721 is low. The findings of immune complex disease are typically reversible when mAb administration stops and the antibody-antigen complexes are cleared from the body.

Based on the phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed.

#### 1.2.5.4 Infections

BOS161721 is expected to diminish the activity of T-cell, B-cell and NK-cell lines. Like other medications modulating immune response, BOS161721 may increase the potential risk for infection, including serious infections. IL-21 produced by CD4+ T-cells is required to sustain the anti-viral function of CD8+ T-cells against chronic viral infections. Nonclinical evidence suggests that the risk of chronic viral infection recurrence or increased severity may occur with IL-21 inhibition.<sup>35</sup>

These conditions will be fully characterized with clinical descriptions and routine laboratory and/or specialty testing and treated where indicated with appropriate local standard of care.

Patients with a history of opportunistic infection, including recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years, or any other underlying pathology predisposing to serious infection, are excluded from studies with BOS161721 (for further details please refer to the current IB for BOS161721).

Patients will be assessed for hepatitis B, and C, and HIV-1/2 combination, at screening.


Cryptosporidium Infection

Cryptosporidium infection was noted in patients with an IL-21 receptor loss-of-function gene mutation and similar findings of cryptosporidium infection have been observed in immunosuppressed liver transplant and human immunodeficiency virus patients. <sup>36,37</sup> Since BOS161721 is expected to diminish the immunosurveillance activity of T-cell, B-cell, and NK-cell lines, a similar risk is biologically plausible with prolonged exposure to BOS161721.

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells,<sup>37</sup> patients with a CD4+ count < 500 cell/mm³ were excluded from the phase 1 SAD study (BOS161721-01). Patients with CD4+ count < 350 cells/mm³ and CD4+ count < 150 cells/mm³ will be excluded from the MAD and POC parts of the study, respectively. Patients exposed to investigational product who develop diarrhea during the course of the study should immediately undergo an assessment for opportunistic infection including stool for ova and parasites and stool examination for cryptosporidium. Positive cryptosporidium in stool sample at screening is an exclusion. Treatment by the Investigator where indicated should be guided by findings and be consistent with local standard of care.

Based on the phase 1 SAD study (BOS161721-01), infections in subjects who received BOS161721 was not observed.

### 1.2.5.5 Malignancy

The stimulatory effect of IL-21 on NK cells and CD8+ T-cells suggests the cytokine may have anti-tumor activity. Nonclinical studies have demonstrated significant anti-tumor effects of IL-21 in a number of tumor models. IL-21 therapy of human metastatic melanoma and renal cell carcinoma has demonstrated POC with significant increases in levels of perforin, granzyme B, and interferon gamma (IFNy) expression in CD8+ T-cells and NK T-cells. Clinical response has been limited in these generally unmanageable diseases.

The impact of treatment with anti-IL-21 therapy on the development or growth of malignancies is not known; however, as with other immunomodulatory biologic agents, treatment with BOS161721 may result in an increase in the risk of malignancies. NK cell suppression by IL-21 neutralization may represent a biological mechanism for a potential risk for malignancy. Patients with a history or current diagnosis of cancer within the past 5 years, with the exception of non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy, are excluded from the study.

Based on the phase 1 SAD study (BOS161721-01), malignancy in subjects who received BOS161721 was not observed.

### 1.2.5.6 Hepatic Function Abnormality

There is no substantial evidence suggesting BOS161721 is associated with liver function abnormality. However, as a precaution, patients with a history of abnormal


alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST > 2 × upper limit of normal [ULN]; total bilirubin > 1.5 × [ULN] and judged by the Investigator to be clinically significant) were excluded from the phase 1 SAD study (BOS161721-01), and will be excluded from this trial. Patients with a positive hepatitis B or C test or a history of alcohol dependence will also be excluded.

Based on the phase 1 SAD study (BOS161721-01), hepatic function abnormality in subjects who received BOS161721 was not observed.

#### 1.2.5.7 Failure of Vaccination

IL-21 is a key cytokine in development of B-cells into immunoglobulin-secreting plasma cells. Abnormal signaling through the IL-21R/Janus Kinase (JAK)3/signal transducer and activator of transcription (STAT3) pathway leads to defective humoral immune responses to both T-dependent and T-independent antigens and impairs the establishment of long-lasting B-cell memory. Abnormal signaling through the pathway has been related to decreased specific antibody responses following vaccination, and to increased susceptibility to encapsulated bacterial infections.<sup>38</sup>

The effect of BOS161721 was evaluated in in vivo single dose studies in Cynomolgus monkey in which the animals received vaccination to T-cell dependent KLH antigen to stimulate a TDAR. These in vivo studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen in a dose-dependent fashion; however, BOS161721 administration did not affect antitetanus toxoid antibody data for IgM, IgG, IgG1, or immunoglobulin E (IgE) during the dosing phase in the same study.

### 1.2.5.8 Potential for Drug-Drug Interactions

Drug-drug interactions were not evaluated in the phase 1 SAD study (BOS161721-01), which included only healthy adult subjects. Use of prescription medications (with the exceptions of oral contraceptives), and over-the-counter (OTC) treatments including herbal supplements such as St John's Wort (except multivitamins), in the 2 weeks prior to screening was prohibited in the SAD study.

See Section 4.5 for other specific exclusion criteria which support lowered risk of interactions, and Section 4.6.1 for corticosteroid (CS) dosing. In addition, Section 1.2.5.6 describes considerations for hepatic function for this study.

### 1.2.5.9 Potential Risk to Fetal Development

No data on preclinical reproductive toxicity are available at the time of this study.

#### 2 STUDY OBJECTIVES AND ENDPOINTS

This trial has separate objectives and endpoints for the MAD phase 1b and POC phase 2 portions of the study. The primary, secondary, and exploratory objectives for each phase, as applicable, are described below with their corresponding endpoints.


BOS161721


## 2.1 Phase 1b Multiple Ascending Dose

| OBJECTIVES | ENDPOINTS |
|---|---|
| Prim | |
| To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of AEs and SAEs, related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness</li> <li>Injection site reactions</li> <li>Columbia Suicide Severity Rating Scale (C-SSRS)</li> <li>12-lead ECGs parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> <li>Clinical laboratory results and change from baseline</li> <li>Physical examinations changes from baseline</li> <li>ADAs</li> <li>Study drug exposure/compliance</li> </ul> |
| Secon | |
| To characterize the PK of<br>BOS161721 and select the optimal<br>dose of BOS161721 based on safety,<br>PK, and PD effects in patients with<br>moderately to severely active SLE | <ul> <li>Pharmacokinetic Endpoints</li> <li>BOS161721 concentration by visit and time point</li> <li>Maximum observed concentration (C<sub>max</sub>), T<sub>max</sub>, area under the concentration-time curve (AUC), terminal elimination half-life (t½), systematic clearance (CL), volume of distribution (V<sub>d</sub>)</li> <li>Pharmacodynamic Endpoints</li> <li>Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype</li> <li>Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit</li> <li>Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit</li> </ul> |
| Explor | |
| • CCI | |




# 2.2 Phase 2 Proof of Concept

| OBJECTIVES | ENDPOINTS |
|---|---|
| Prim | nary |
| To demonstrate a superior effect of<br>BOS161721 at the chosen dose<br>compared with placebo for response<br>on the SRI-4 | <ul> <li>Primary Efficacy Endpoint</li> <li>The proportion of patients with a SRI-4 response at Day 210 (see Section 6.3.4.1)</li> </ul> |
| Secon | ndary |
| To demonstrate a superior effect of<br>BOS161721 at the chosen dose<br>compared with placebo for response<br>on clinical indicators of SLE activity, in<br>adult patients with moderately to<br>severely active SLE on limited<br>background standard of care<br>treatment | <ul> <li>The proportion of patients with: <ul> <li>SRI-4 response at each visit</li> <li>SRI-5 and SRI-6 response at each visit (Section 6.3.4.2)</li> <li>a sustained reduction from baseline of oral corticosteroid (CS) (≤ 7.5 mg/day and &lt; Day 0 dose) between Day 150 and Day 210</li> <li>new or recurrent BILAG flares (≥ 1 qualifying BILAG A or &gt; 1 qualifying BILAG B) through Day 210</li> <li>PGA worsening</li> <li>a BICLA response</li> <li>a CLASI response</li> </ul> </li> </ul> |


- medication failures The changes and percent changes from baseline in:
  - **CLASI**
  - **PGA**
  - Total number of swollen joints, tender joints, and active joints (swelling and tenderness in the same joint) in the ACR-28 joint count
  - SLEDAI-2K
  - SLICC/ACR damage index
- Time to medication failure
- Group mean percent reduction in CS administration from baseline Day 0 dose through Day 210 in patients receiving ≥ 7.5 mg/day prednisone equivalent at Day 0
- Duration of longest SRI-4 response
- Time to first BILAG flare (≥ 1 new or recurrent BILAG A or > 1 new or recurrent BILAG B) relative to baseline through Day 210

#### Safety

To assess safety and tolerability of repeat doses of BOS161721 at the chosen dose administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment

#### Safety Endpoints

- Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness
- Injection site reactions
- C-SSRS
- 12-lead ECGs parameter results at each visit and change from baseline
- Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline
- Clinical laboratory results and change from baseline
- Physical examinations changes from baseline
- **ADAs**
- Study drug exposure/compliance






### 3 STUDY PLAN

### 3.1 Study Design

This is a phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, eligible patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly.

The trial will consist of 2 double-blinded portions: MAD phase 1b and POC phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

SLE disease activity assessment data will be centrally reviewed by medical monitor and sponsor to ensure the scores are clinically meaningful and compliant with specific definition. The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease activity. Further details on the content and methods of data reports by the medical monitor and sponsor will be outlined in the Medical Data Review Plan along with the processes and procedures that will be followed.

### 3.1.1 Multiple Ascending Dose Phase 1b

The MAD portion will consist of 3 cohorts:

- Cohort 1 (20 mg SC) will include 6 patients
  - 5 patients will receive BOS161721 (active group) and 1 patient will receive placebo (placebo group)
- Cohorts 2 (60 mg SC) and 3 (120 mg SC) will include 12 patients each
  - 9 patients in the active group and 3 in the placebo group


Doses selected for each of the 3 cohorts is based on a 90 day safety, tolerability, PK and PD data review from the phase 1 SAD study (BOS161721-01) in healthy subjects. All doses selected for the MAD part of the study are projected not to exceed the mean exposure of that achieved at the highest dose in the SAD study.

#### 3.1.1.1 Dose Escalation for the MAD Portion

The MAD portion of the study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after the DMC evaluation of the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after the DMC evaluation of the safety and tolerability data from Cohorts 1 and 2. Each cohort will continue at their assigned dose level through their respective 6-month treatment periods (see Study Schematic, Section 3.3). If patients discontinue the study in a cohort prior to adequate safety follow-up, he/she may be replaced.

Criteria for dose escalation are further described in the DMC Charter. See Section 3.1.1.2 for additional details about DLTs.

### 3.1.1.2 Dose Limiting Toxicity (DLT)

Severity of adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs occurring after study drug administration, which are attributable to the study drug, will be considered DLTs:

#### Hematologic:

- Grade 4 neutropenia
- Grade 3 neutropenic infection
- Grade 3 thrombocytopenia with bleeding
- Grade 4 thrombocytopenia

#### Non-Hematologic:

- Grade 3 or above toxicities, persisting after optimal treatment with standard medical therapy (e.g., anti-emetics, anti-diarrheals)
- Drug-induced liver injury ([DILI], Hy's Law), as defined in Section 6.2.2.6.3 Investigators should always manage their patients according to their medical judgment which may include interruption of study drug based on the particular clinical circumstances.


#### 3.1.1.3 DMC Recommendations

During scheduled meetings, the DMC will review relevant study data for safety or benefit-risk concern. During the MAD part of the study, the DMC may provide the following recommendations to the sponsor:

- Expanding a cohort at a specific dosing level, or repeating a lower dose in a subsequent cohort
- Continuing a dose level for a given cohort
- Escalating a dose level for a subsequent cohort
- Termination of current or previous cohort(s)

Further dosing in a given cohort will be halted if 2 or more DLTs are identified intra- and inter-patients dosed. For the POC portion, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC phase 2 part of the study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD portion. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available 30 days after the last patient from Cohort 3 receives the third dose. Details are provided in the DMC Charter.

#### 3.1.2 POC Phase 2

#### 3.1.2.1 BOS161721 POC Dose Selection and Justification

The dose for the POC portion of the study is 120 mg administered SC monthly (a total of 7 doses). The rationale for the BOS161721-02 phase 2 POC dose selection was based on cumulative safety, tolerability, immunogenicity, PK, and PD data available from an interim analysis (IA) performed during the MAD phase 1b portion of the trial.

The data cut-off for this IA occurred on CCI and and included all 6 patients and 7 doses from Cohort 1 (20 mg), 12 patients and 6 doses from Cohort 2 (60 mg), and 12 patients and 4 doses from Cohort 3 (120 mg).

The safety analysis focused on incidence and severity of all AEs, SAEs, and predetermined adverse events of special interest (see Section 6.2.2.6). The DMC and designated unblinded Boston Pharmaceuticals team met on CCI and and did not identify any untoward safety signals at any BOS161721 dose levels.

Because there were no safety, tolerability, or immunogenicity trends observed at the time of the IA, the phase 2 POC dose selection was made based on available PK and PD data. pSTAT3 levels were assessed as the primary PD biomarker of IL-21R signaling levels. This is because IL-21R signaling, upon IL-21 binding, initially involves phosphorylation of JAK1/JAK3 which dissociate from the receptor complex, and phosphorylate STAT3 which translocates to the nucleus and drives IL-21-regulated gene expression.


CCI



The 120 mg dose was communicated to site Investigators participating in the POC phase 2 portion, and to Institutional Review Boards (IRBs) and the Independent Ethics Committee (IEC).

### 3.1.2.2 POC Study Design

For the POC part of the study, approximately 110 additional patients will be randomized to active or placebo groups in a 2:1 ratio.

As in the MAD part of the study, each patient in the POC portion may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Table 1 and Table 4).

DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.

### 3.2 Randomization and Blinding

This is a randomized, double-blind study.

Patients meeting all inclusion and exclusion criteria will be centrally randomized to either placebo or BOS161721 using an IWRS according to a randomization list generated by an independent, non-study statistician. Randomization will be performed separately for each study portion and separately for each cohort in the phase 1b and 2 portions as follows:

| Phase/Cohort | Number of Patients | Randomization Ratio BOS161721:Placebo |
|---|---|---|
| Phase 1b/Cohort 1 | 6 | 5:1 |
| Phase 1b/Cohort 2 | 12 | 3:1 |
| Phase 1b/Cohort 3 | 12 | 3:1 |
| Phase 2 | Approximately 110 | 2:1 |

<sup>\*</sup>Additional patients may be enrolled to ensure sufficient numbers of patients are in the full analysis set (FAS).

Eligible patients will be assigned to the study portion which is active at time of enrollment. Similarly, patients in the phase 1b MAD will be assigned to the cohort which is active. Each patient will be assigned a unique randomization number which will not be reused.

All patients, Investigators, and study team participants will be blinded to treatment assignment. An independent biostatistician not otherwise involved on the study will be unblinded and prepare materials for the IA, ad hoc analyses as needed, and the DMC


safety reviews. The DMC will review unblinded data during safety reviews and the IA. A limited team at Boston Pharmaceuticals will review unblinded results from the phase 1b MAD portion during the IA to determine the dose that will be used for the phase 2 POC portion of the study. Details regarding maintenance of the blinding and content of data reviews will be described in the DMC charter or related study documentation.


### 3.3 Study Schematic

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2



A = active drug (BOS161721); P = placebo


BOS161721 Boston Pharmaceuticals, Inc


#### 3.4 Schedule of Assessments

Table 1. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | Tr | eatmen | t Period | Follow- | up | | | Safe | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28 to -1 | 0 | 15<br>(± 3) | 30<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187 <sup>b</sup><br>(± 3) | 195 <sup>b</sup><br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| GENERAL ASSESSMENTS | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | Χ | | | | | | | | | | | | | |
| Medical history | Х | | | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | | | |
| SLICC Criteria for SLE | Χ | | | | | | | | | | | | | |
| Concomitant medication <sup>c</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Randomizationd | | Х | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | х | | Х | Х | Х | х | х | Х | | | | | |
| | SAFETY ASSESSMENTS | | | | | | | | | | | | | |
| Full physical exam | Х | Х | | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Screening assessments will be performed over more than 1 visit.


<sup>&</sup>lt;sup>b</sup> PK samples will only be collected at the investigational sites that participate in the PK portion of the study. On PK only days (i.e., Day 187 and Day 195 when no laboratory assessments are scheduled) samples will be collected at the investigational sites of the selected countries that participate in the PK portion of the study. Patients not participating in PK are not required to return for investigation site visits on Days 187 and 195.

<sup>&</sup>lt;sup>c</sup> Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the dose must be stable for at least 6 weeks prior to Day 0 (randomization day). See Section 4.6.1 for further details.

<sup>&</sup>lt;sup>d</sup> Randomization should occur after patient eligibility has been confirmed. The actual randomization procedure can be completed on Day -1 after eligibility confirmation or the morning of Day 0 prior to dosing for logistical purposes.

BOS161721 Boston Pharmaceuticals, Inc

Clinical Study Protocol: BOS161721-02


Table 1. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | Tre | eatmen | t Period | Follow- | up | | | Safe | ty Follo | ow-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28 to -1 | 0 | 15<br>(± 3) | 30<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187 <sup>b</sup><br>(± 3) | 195 <sup>b</sup><br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| Chest x-ray <sup>e</sup> | X | | | | | | | | | | | | | |
| C-SSRS | Х | Х | | | | Х | | | Х | | | | | |
| AEs and SAEs | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ |
| 12-lead ECG <sup>f</sup> | Х | Х | | Х | | Х | | | | | | | | Χ |
| Injection site reaction assessment | | Χg | | Х | Х | Х | Х | Х | Х | Х | х | Х | Х | Х |
| Targeted physical examination | | | Х | Х | Х | Х | х | х | Х | | | Х | Х | Х |
| Vital signs (BP, HR, and temperature) <sup>h</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | Х | Х | Х |
| | | | E | FFICAC | Y ASSI | SSME | NTS | | | | | | | |
| BILAG-2004 Index | Х | Х | | Х | Χ | Х | Х | Х | Х | | | Х | Х | Χ |


e If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0)

f ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws

<sup>&</sup>lt;sup>9</sup> Injection site reaction assessments to be performed at 2 hours postdose

<sup>&</sup>lt;sup>h</sup> Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours (± 15 minutes) postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 187 and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection

BOS161721 Boston Pharmaceuticals, Inc


Table 1. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | Tre | eatmen | t Period | Follow- | up | | | Safe | ty Follo | ow-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28 to -1 | 0 | 15<br>(± 3) | 30<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187 <sup>b</sup><br>(± 3) | 195 <sup>b</sup><br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| SLEDAI-2K | Χ | Xi | | Х | Χ | Х | Χ | Χ | Х | | | Х | Х | X |
| PGA | Χ | Χ | | Χ | Χ | Χ | X | Χ | X | | | Х | X | X |
| ACR-28 joint count | Х | Х | | Х | Х | Х | Х | Х | Х | | | Х | Х | Х |
| CLASI | Х | Х | | Х | Х | Х | Х | Х | Х | | | Х | Χ | Х |
| CCI | | Х | | Х | Х | Х | Х | Х | Х | | | Х | Χ | Х |
| SLICC/ACR Damage Index | | Х | | | | | | | Х | | | | | |
| CCI | | Х | | Х | Х | Х | Х | Х | Х | | | Х | Х | Х |
| | | | LAE | ORAT | ORY AS | SESSN | IENTS | | | • | | | • | |
| CD4+ count | Х | Х | Х | Х | | Х | | | Х | | | | | |
| Clinical laboratory<br>assessments (hematology<br>and clinical chemistry) <sup>j</sup> | X | х | | Х | х | Х | x | Х | Х | | | Х | Х | Х |
| Coomb's test direct <sup>k</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | Х | X | | X | | | X | | | | | |
| Plasma CCI | X | X | | X | Х | X | Х | Х | X | | | Х | Х | Х |
| Plasma CCI & | | X | Х | Х | | Х | | | Х | | | | | |


<sup>&</sup>lt;sup>1</sup> SLEDAI-2K should be done before randomization and dosing on Day 0 as SLEDAI-2K < 6 is exclusionary

<sup>&</sup>lt;sup>j</sup> Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting

<sup>&</sup>lt;sup>k</sup> When clinically indicated for hemolytic anemia

BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02


Table 1. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | Tre | eatmen | t Period | Follow- | up | | | Safety Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28 to -1 | 0 | 15<br>(± 3) | 30<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187 <sup>b</sup><br>(± 3) | 195 <sup>b</sup><br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| ADA <sup>I</sup> | | Χ | X | Χ | Χ | X | | | Χ | | | | | Χ |
| nAb <sup>m</sup> | | | | | | Х | | | X | | | | | |
| CCI | | Х | Х | | | Х | | | Х | | | | | Х |
| CCI | | Х | | | | | | | | | | | | |
| CCI | x | x | | X | × | X | x | x | X | | | Xn | Xn | Xn |
| CRP | Х | | | | | Х | | | | | | | | Х |
| Serum pregnancy test (women) | Х | | | | | | | | | | | | | |
| FSH (postmenopausal women) | Х | | | | | | | | | | | | | |
| Urine pregnancy test (women)º | | Х | | Х | Х | Х | Х | х | Х | | | | | Х |
| TB test (QuantiFERON®-TB Gold In-Tube)® | Х | | | | | | | | | | | | | |
| Serology (hepatitis B and C, HIV-1/2 combination) | Х | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed (analyzed) if the patient had a positive ADA on Day 90


<sup>&</sup>lt;sup>m</sup> nAb is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90

will not be analyzed during safety follow-up visits

<sup>°</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits

BOS161721

Clinical Study Protocol: BOS161721-02


Table 1. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screen | Enroll | | | Tr | eatmen | t Period | Follow- | up | | | Safety Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | -28 to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| Stool sample <sup>p</sup> | X | | | | | | | | | | | | | |
| Spot urine for protein/creatinine ratio | x | х | | Х | Х | Х | x | х | Х | | | Х | Х | х |
| Urinalysis | Х | Χ | | Χ | Χ | Χ | Х | Х | Х | | | Х | Х | Χ |
| | PK Labs <sup>b</sup> | | | | | | | | | | | | | |
| Predose | | Х | | Х | Х | Х | Х | Х | Х | | | | | |
| Postdose | | | Х | | | | | | | Х | Х | Χ | Х | Х |

Abbreviations: ACR = American College of Rheumatology; ADA = anti-drug antibody; AE = adverse event; College of Rheumatology; ADA = anti-drug antibody; AE = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; College of Rheumatology; FSH = follicle stimulating hormone; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; SAE = serious adverse event; College of Rheumatology; ADA = anti-drug antibody; AE = adverse event; College of AEA = adve


P Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium

### 3.5 End of Study

**End of Study (Individual Patient)**: A patient is considered at the end of study if he/she has withdrawn, prematurely discontinued, or completed all of the study procedures including the last visit.

**End of Study (End of trial):** The end of the study is defined as the date of the last visit of the last patient in the study globally, or the date of which the last patient withdraws or discontinues if all prior enrolled patients have already completed/withdrawn.

### 4 POPULATION

### 4.1 Participant Recruitment

Advertisements approved by the IRB, and Investigator databases, may be used as recruitment procedures for adult men and women with moderately to severely active SLE.

#### 4.2 Number of Patients

Approximately 140 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD phase 1b portion, and approximately 110 additional patients will be randomized in the POC phase 2 portion. Note that approximately 14 dropouts are assumed in the POC phase 2 portion.

### 4.3 Patient Screening

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Table 1 and Table 4]) for this study must be performed between Day -28 and Day -1.

#### 4.4 Inclusion Criteria

Patients who meet the following criteria will be considered eligible to participate in this clinical study:

1. Men and women, ages 18 to 70 years, inclusive.


2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.

- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion or Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously.
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA ≥ 1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
- 5. At screening, the total SLEDAI-2K score must be ≥ 8, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.
- 6. A clinical SLEDAI-2K score of ≥ 6 at screening at Day 0. Clinical SLEDAI-2K score is defined as follows:
  - a. Contains points from arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, or vasculitis
  - b. Excludes parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement. thrombocytopenia, and leukopenia

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

- 7. Patients must have at least 1 qualifying A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system. If a BILAG B score is due to BILAG number 6, mild skin eruption, the CLASI activity score including erythema and scale/hypertrophy must be ≥ 3 excluding points from mucosal ulcers and alopecia.
  - BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis defined by BOTH swelling and tenderness in ≥ 6 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living (ADLs) that has been present on several days


( > 4 days) cumulatively over the past 30 days, including at the time of the screening visit. See Appendix 5 for additional detailed specifications.

- Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):
  - Ambulation, toileting, grooming- including bathing and dressing; feeding oneself
- ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis defined by BOTH swelling and tenderness in ≥ 3 joints, (observed or through patient history), with some loss of functional range of movements manifested by effects on instrumental ADLs such as:
  - Cooking, driving, using the telephone or computer, shopping, cleaning, etc., and has been present on several days over the last 30 days, and is present at the time of the screening visit

Note: Hips, shoulders, back, neck, and temporomandibular joints do not count towards the total number of joints with active synovitis.

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in at least 1 other body system for a total of 2 "B" BILAG body system scores.

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to Day 0) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. If AZA, myocophenolate mofetil, mycophenolic acid, hydroxychloroquine, or MTX were discontinued prior to screening, the washout period must be ≥ 12 weeks
  - c. Corticosteroids (prednisone or prednisone-equivalent) at a stable dose of up to 30 mg/day for at least 6 weeks prior to Day 0 (see Appendix 3)
    - i. For patients whose only SLE treatment is CS, the stable CS dose must be ≥ 10 mg/day for at least 6 weeks prior to Day 0 and no more than 30 mg/day at the time of randomization
    - ii. Topical steroids may be used, but the dose must be stable for at least 6 weeks prior to Day 0. PRN topical steroids are not permitted
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding


c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks.

- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks.
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures.

#### 4.5 Exclusion Criteria

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE.
- 2. Other systemic autoimmune disease (e.g., erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic sclerosis, or vasculitis not related to SLE).
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study.
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed.
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed.
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS.
- 7. Concomitant illness that, in the opinion of the Investigator or the sponsor or their designee, is likely to require additional systemic glucocorticosteroid therapy during the study, (e.g., asthma), is exclusionary.
  - a. However, treatment for asthma with inhalational CS therapy is allowed.


- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study. (See Section 4.6.2 for prohibited concomitant medication).
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization.
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years.
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
- 12. Cryptosporidium in the stool sample at screening.
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening.
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening.
- 15. CD4+ count < 150/μL at screening.
- 16. Platelets < 50,000/mm³ ( $50 \times 10^9$ /L) or < 35,000/mm³ ( $35 \times 10^9$ /L) if related to SLE, at screening.
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if related to SLE.
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol).
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 mL/minute based on Cockcroft-Gault calculation<sup>39</sup>:
  - GFR = ([1 for male] or [0.85 for female])  $\times$  (140 Age)  $\times$  BW/(72  $\times$  Creatinine).
- 20. Serum ALT and/or serum AST > 2 × ULN at screening, unless explicitly related to lupus based on the Investigator's judgment.
- 21. Creatinine kinase (CK) > 3.0 × ULN at screening, unless it is related to lupus myositis.
- 22. Total bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome).
- 23. Any other laboratory test results that, in the opinion of the Investigator or the sponsor or sponsor's designee, might place a patient at unacceptable risk for participating in this study.


24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (e.g., IgG protein) or molecules made of components of

monoclonal antibodies.

25. History substance and/or alcohol abuse or dependence within the past 1 year, at the Investigator's judgment.

- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer *in situ* resolved by excision).
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (e.g., cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, sponsor or sponsor's designee, would make the patient inappropriate for entry into this study.
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial.
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer.
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4 or 5 on the C-SSRS.
- 31. Current or pending incarceration.
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
- 33. Currently taking a total daily dose of > 30 mg morphine or morphine equivalent (see Appendix 7).
- 34. Body mass index (BMI)  $\geq$  40.0.

#### 4.6 Concomitant Medications

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Patients should stay on stable regimen (not PRN) of other concomitant medications for the treatment of SLE (e.g., analgesics, nonsteroidal anti-inflammatory drugs [NSAIDs], statins, ACE inhibitors/ARBs and other antihypertensive drugs), unless changes in these treatments are clinically indicated. Patients should refrain from Tylenol, NSAIDs, and any pain medications including tramadol and other opiates for at least 12 hours before each visit, with the exception of the Screening Visit.


Use of any other drugs for non-SLE conditions, including over-the-counter medications and herbal preparations, should remain stable unless change or addition is clinically necessary. Discussion with the medical monitor prior to initiation of new medication is strongly recommended. Any concomitant therapies must be recorded on the eCRF. Prior and concomitant medication use will be recorded for the 30 days prior to screening until the last follow-up visit. In addition, historical treatment for SLE (including immunosuppressant, anti-malarial, corticosteroid, and/or biologic agent including investigational agents) will be recorded for the 48 weeks prior to screening in the eCRF.

#### 4.6.1 Corticosteroid

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the Investigator's clinical judgment and best standard of care. See Appendix 3 for examples of equivalents.

- A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study. For patients whose only SLE treatment is steroids, their stable steroid dose must be at least 10 mg/day and no more than 30 mg/day for a minimum of 6 weeks at time of randomization on Day 0
- Topical steroids may be used, but the dose must be stable for at least 6 weeks prior to Day 0, and be maintained at a constant dose throughout the study duration until the rashes resolve. PRN topical steroids are not permitted
- Once the patient has received the first dose of study drug (Day 0), tapering of oral steroids will be highly encouraged and should be continually evaluated during the protocol-allowed tapering windows (Day 0 through Day 150) with the target of achieving a CS daily dose of < 7.5 mg and < Day 0 dose between Day 150 and Day 210
- Between Day 150 and Day 210 (i.e., within 60 days of primary endpoint assessments), oral CS doses must be held constant
- CS Burst for SLE-related Indications
  - After Day 0 (first dose of study drug), a maximum of 1 oral CS "burst" equivalent to ≤ 40 mg/day prednisone for increased SLE disease activity will be allowed between Day 0 and Day 120, which must be tapered down to the baseline (Day 0) CS dose or lower within 14 days of initiation of the "burst". Any "burst" continuing after Day 120 or occurring after Day 120 is considered a protocol deviation.
  - Alternatively, a single intramuscular (IM) dose of methylprednisolone ( < 40 mg) is permitted during this period</li>

CS Burst for Non-SLE-related Indications.

A single treatment of oral prednisone equivalent of  $\leq$  40 mg/day for 14 days is permitted for a non-SLE indication, though it must be completed prior to Day 120. No long acting steroid injections are permitted.

Note: Treatment with inhaled CS are allowed for the treatment of non-SLE-related indications only (e.g., for asthma).


Any other increase from baseline of CS dose or systemic use of CS of any kind (including intra-articular and intravenous administration) are not permitted from Day 0 through Day 210 and will result in the patient being considered a treatment failure. There is no restriction of CS usage after Day 210.

#### 4.6.2 Other Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in Appendix 4. All medications taken within 30 days prior to screening must be recorded on the eCRF.

- 1. Prior exposure to BOS161721
- 2. Patients who have received treatment with anti-CD20 monoclonal antibodies within 24 weeks of screening
- 3. Patients who have received treatment with cyclophosphamide within the 24 weeks prior to screening
- 4. Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria within 4 weeks for oral use or 8 weeks for topical use of screening
- Patients who are currently receiving or are scheduled to receive plasmapheresis or lymphapheresis therapy, or have received such therapy within 24 weeks prior to screening
- 6. Patients who have received any live vaccines within 30 days of screening. Note: Furthermore, live vaccines should not be used during the course of the study and within the 2 months following last dose. Other inactivated vaccines such as tetanus, etc., may be used according to local guidelines during treatment period
- 7. Patients who are scheduled or anticipated to have elective surgery during the course of the study
- 8. Initiation of new immunosuppressant or anti-malarial agent is not permitted. Note: Dose reduction or replacement may be allowed due to intolerability or shortage for patients on a stable dose prior to study initiation

## 4.7 Women of Childbearing Potential

WOCBP is defined as any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) and is not postmenopausal.


See Section 4.7.2 for detailed information regarding contraceptive requirements for WOCBP.

#### 4.7.1 Determination of Menopause

Menopause is defined as at least 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes. Women under the age of 55 years must have a documented serum FSH level > 40 mIU/mL at screening to confirm menopause.

### 4.7.2 Contraception

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks, due to the mean terminal  $\frac{1}{2}$  life of the study drug.

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks, due to the mean terminal ½ life of the study drug.

Investigators shall counsel WOCBP and men who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and men who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

- Patients must agree to either complete abstinence, defined as a complete avoidance of heterosexual activity, or the use of 2 methods of effective contraception from the following:
- Male condoms with spermicide
- Diaphragm with spermicide
- Cervical cap with spermicide
- Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, patches and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
- IUDs, such as ParaGard<sup>®</sup>
- Vasectomy
- Note: Women who are abstinent while participating in the study must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the patient chooses to forego complete abstinence


 Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing

#### 4.8 Deviation from Inclusion/Exclusion Criteria

Deviation from the inclusion or exclusion criteria will not be allowed. If deviation of inclusion/exclusion criteria is discovered after randomization, the Investigator should contact the medical monitor for discussion. A decision will be made whether to allow a patient to continue or withdrawal from the study medication.

See Section 6.8 for additional details.

### 4.8.1 Patient Withdrawal and Replacement

See Section 5.5 for reasons for removal from the trial. Withdrawn patients may be replaced during the MAD part of the study after discussion between the Principal Investigator or designee and sponsor.

#### 5 STUDY PROCEDURES

Refer to the eCRF completion guidelines for data collection requirements and documentation of study assessments/procedures.

### 5.1 Screening

Screening will be the same for both the MAD and POC portions of the study.

Screening will take place from Day -28 to Day -1, and assessments may be performed over more than 1 visit. Confirmation that the most current IRB/IEC approved informed consent form (ICF) has been signed must occur before any study-specific screening procedures are performed. Procedures that are part of standard of care are not considered study-specific procedures and may be performed prior to informed consent and used to determine eligibility.

All screened patients will be assigned a unique screening number. The screening number will include a 3-digit site number and a 4-digit sequential number to identify patients from the time of screening. Only eligible patients who are confirmed by central review as meeting the inclusion/exclusion criteria, listed in Section 4.4 and Section 4.5 respectively, will be enrolled in the study. Screened patients who drop out of the clinical study before randomization will be recorded as screen failures. If rescreening occurs, the site will assign a new screening number.

Specific procedures at the screening visit will include:

- Medical history documentation
- Review of inclusion and exclusion criteria


- Patient medical records must contain documentation of SLE diagnosis
- C-SSRS
- Concomitant medication documentation
- Demographics
- Full physical examination
- Vital signs
- Chest x-ray (a prior x-ray can be used if taken within 12 weeks of screening date)
- Laboratory evaluations (non-fasting):
  - Hematology and clinical chemistry
  - Serology (Hepatitis B and C; HIV-1/2 combination)
  - o TB test
  - o CRP
  - Direct Coomb's test (if indicated for hemolytic anemia)
  - CD4+ count, total IgG and IgM levels, plasma CO
  - Serum pregnancy test (WOCBP)
  - FSH (postmenopausal women under age 55 years)
  - Spot urine for protein/creatinine ratio
  - Urinalysis
  - o Stool sample
- 12-lead ECG
- SLE-related indices [BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, Physician's Global Assessment (PGA) of disease activity]
- Screening procedures are listed in the Schedule of Assessments (Table 1 and Table 4), and details are provided in Section 6.

#### 5.1.1 Retesting During Screening Period

A single retesting of laboratory parameters and/or other assessments during the screening period is permitted (in addition to any parameters that require a confirmatory value) only if:

- medically indicated
- there is evidence a laboratory sample was mislabeled, indeterminate, inadequately processed, and/or deteriorated in transit to the central laboratory

Any new result will override the previous result (i.e., the most current result prior to randomization) and is the value by which study inclusion/exclusion will be assessed, as it represents the patient's most current clinical state. This will also apply to patients who are being rescreened.


### 5.2 Enrollment/Randomization and Day 0 Treatment

Randomization should occur after patient eligibility for enrollment has been confirmed by the central eligibility review. The central eligibility review team has the final decision on patient eligibility and can decide the patient is not eligible for the study based on their review of the eligibility packet.

Prior to randomization, the study site should confirm that the patient still meets inclusion/exclusion criteria (especially SLE disease activity and treatment). The site will obtain a randomization number when registering the patient in interactive web response system (IWRS). All patients will receive BOS161721 or placebo according to the kit number assigned by the IWRS randomization scheme.

After randomization, procedures include:

- PROs: CCI
- C-SSRS
- Laboratory evaluations (fasting):
  - Hematology and clinical chemistry
  - Direct Coomb's test (if indicated for hemolytic anemia)
  - CD4+ count, total IgG and IgM levels, plasma cci , plasma cci and , whole blood for leukocyte immunophenotype (leukocyte immunophenotype for MAD patients only)
  - o ADA
  - pSTAT3 (predose [trough] samples only in phase 1b)
  - o CCI
  - See Table 4 and Table 1 for details of PK sampling in the MAD and POC portions
  - Urine pregnancy test will be collected on WOCBP prior to study drug administration
  - Spot urine for protein/creatinine ratio
  - o Urinalysis
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Full physical examination
- Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours [± 15 minutes] postdose on Day 0)
- 12-lead ECG (prior to PK blood draw)
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, PGA)


- SLICC/ACR damage index
- Study drug administration:

BOS161721

- Administration of BOS161721 or placebo will take place on-site, and is discussed in Section 7.3.
- Injection site reaction assessment performed at 2 hours postdose

Procedures on Day 0 are listed in the Schedule of Assessments (Table 1 and Table 4), and details are provided in Section 6.

All patients who are enrolled, randomized, and receive study drug, or undergo study-specific procedures should reconsent with any updated versions of IRB/IEC approved informed consents during study participation as applicable and per institutional guidelines.

### 5.3 Treatment Period/Follow-Up Visits

The following procedures will be performed as indicated in the Schedule of Assessments (Table 1 and Table 4). See Schedule of Assessment tables for allowable windows for each visit.

- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- PROs: CC
- Urine pregnancy tests will be collected on WOCBP prior to study drug administration
- Injection site reaction assessments will be performed predose
- Direct Coomb's test (if indicated for hemolytic anemia)
- Spot urine for protein to creatinine ratio
- Urinalysis
- CCI
- Plasma CCI
- PGA, BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, and the CLASI will be completed
- SLICC/ACR Damage Index will be completed at Day 180
- C-SSRS
- ECGs prior to PK blood draw
- See Table 4 and Table 1 for details of PK sampling in the MAD and POC studies, respectively
- Fasting hematology and chemistry assessments
- The CD4+ count and total IgG and IgM levels


- Plasma column and column, ADA, and whole blood for leukocyte immunophenotype (leukocyte immunophenotype for MAD patients only)
- pSTAT3 (predose [trough] samples only phase 1b)
- nAb will be analyzed by central lab if patient is positive for ADA
- CRP
- CCI

### 5.4 Safety Follow-Up Visits

Safety follow-up visits will take place at Days 210, 240, and 270. These visits will include the following assessments as indicated in the Schedule of Assessments (Table 1 and Table 4):

- PROs: CCI
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Injection site reactions
- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Spot urine for protein/creatinine ratio and urinalysis
- Concomitant medication documentation
- BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, and PGA
- Fasting clinical laboratory assessments (hematology and clinical chemistry)
- Direct Coomb's test (if indicated for hemolytic anemia)
- Plasma CCI
- CCI
- 12-lead ECG (prior to PK blood draw)
- CRP
- ADA
- CCI
- Urine pregnancy test
- See Table 1 and Table 4 for details of PK sampling in the MAD and POC portions, respectively

#### 5.5 Premature Discontinuation

While patients are encouraged to complete all study evaluations, they may withdraw from the study at any time and for any reason. Every effort will be made to determine why any patient withdraws from the study prematurely. If the patient is unreachable by telephone, a registered letter, at the minimum, should be sent to the patient requesting him/her to contact the clinic.


All patients who withdraw from the study with an ongoing AE or SAE must be followed until the end of study or until the event is resolved or deemed stable, respectively.

If a patient withdraws prematurely after dosing, an end of treatment (EOT) visit should be performed (Day 180) and a last follow-up visit 90 days after dosing should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 5.4).

Patient participation may be terminated prior to completing the study and the reason recorded as follows:

- AF/SAF
- Protocol deviation
- Lost to follow-up
- Patient withdraws consent at their own request
- Investigator decision
- Decision by the sponsor (other than AE/SAE, protocol deviation, or lost to follow-up) Withdrawn patients may be replaced after discussion between the Investigator or designee and sponsor.

#### **Contingency Plans During the COVID-19 Pandemic** 5.6

- Safety oversight: In case a patient cannot return to the study site for the scheduled visit, the site staff will contact the patient remotely for safety follow up, for example, via telephone or video conferencing.
- Central Laboratory: In the case there are courier issues that will prevent the protocol-required laboratory specimens to be sent to the study core laboratory. the site should have the safety laboratory speciments (Table 2: Hematology, Chemistry, and Urinalysis) sent to their local laboratory for analysis and review by the study physician.
- Investigational Product Dosing: In cases when dosing cannot be performed during the protocol-designated windows, the Investigator should discuss each case with the Sponsor to determine whether it is a missed visit or whether the dosing can be performed outside protocol windows (as a protocol deviation). A minimum of 2 weeks must be maintained between consecutive doses. Patients who miss more than 2 doses of the study drug (whether consecutive or not) will be discontinued from the study and will undergo assessments as outlined in Section 5.5 (Premature Discontinuation).


#### **6 ASSESSMENTS**

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances, outside of the control of the Investigator, which may make it unfeasible to perform the test. In these cases, the Investigator will take all steps necessary to ensure the safety and wellbeing of the patient. When a protocol required test cannot be performed the Investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. All protocol violations are entered directly into the eCRFs.

### 6.1 Medical History, Demographic and Other Baseline Information

The medical history comprises:

- General medical history
- Documentation of SLE diagnosis
- Historical medication therapy for SLE

The following demographic information will be recorded:

- Age
- Ethnic origin (Hispanic/Latino or not Hispanic/not Latino)
- Race (White, American Indian/Alaska Native, Asian, Native Hawaiian or other Pacific Islander, Black/African American)
- Height (without shoes, in cm)
- Body weight, without shoes (kg)
- BMI [kg/m²]

Other baseline characteristics will be recorded as follows:

- Concomitant medication documentation (see Section 4.6)
- Status of child bearing potential and contraception

### 6.2 Safety Assessments

### 6.2.1 Laboratory Assessments

Laboratory tests will be performed at times defined in the Schedule of Assessments (Table 1 and Table 4). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

A central laboratory will be used (with the exception of urine pregnancy tests) to ensure accuracy and consistency in test results. Laboratory/analyte results that could unblind the study (i.e., biomarker results) will not be reported to investigative sites. Urinalysis


will be performed on midstream, clean catch specimens. Some biomarkers listed above will not be drawn at some sites due to geographical logistical challenges. See the laboratory manual for details.

Endpoint analyses will be based on changes from baseline assessments at Days 120 and 210.

**Table 2. Laboratory Tests** 

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| Hemoglobin Hematocrit RBC count RDW MCV MCH MCHC Platelet count WBC count CD4+ count Total neutrophils (Abs) Eosinophils (Abs) Monocytes (Abs) Basophils (Abs) Lymphocytes (Abs) | BUN Creatinine Glucose (fasting) Calcium Sodium Potassium Chloride Total CO <sub>2</sub> (bicarbonate) AST, ALT Total bilirubin Alkaline phosphatase Creatine kinase Uric acid Albumin Total cholesterol (fasting) LDL-C (fasting) HDL-C (fasting) Triglycerides (fasting) Total protein PT/INR | pH Glucose (qual) Protein (qual) Blood (qual) Ketones Nitrites Leukocyte esterase Urobilinogen Urine bilirubin Microscopy <sup>a</sup> | Spot urine for protein/creatinine ratio FSHb Urine pregnancy testc QuantiFERON®-TB Gold In-Tube test (QFT-G)d Serologyd (Hepatitis B and C; HIV-1/2 combination) Stool samplec Serum pregnancy test |
| | Additional Testsf (potential Hy's Law) AST, ALT (repeat) Total bilirubin (repeat) Albumin (repeat) Alkaline phosphatase (repeat) Direct bilirubin Indirect bilirubin GGT Prothrombin time/international normalized ratio (repeat) Creatine kinase (repeat) | | Immunogenicity, PD and other Biomarker Tests ADA nAb <sup>9</sup> pSTAT3 (predose [trough] samples only in phase 1b) Total IgG & IgM Plasma CCI Plasma CCI Plasma CCI Whole blood for leukocyte immunophenotype (for MAD patients only) CCI C |


**Table 2. Laboratory Tests** 

Hematology Chemistry **Urinalysis Other Safety Tests** Abbreviations: Abs = absolute; ADA = anti-drug antibody; ALT = alanine aminotransferase; ; AST = aspartate aminotransferase; BUN = blood urea nitrogen; C = complement; CD4+ = cluster of differentiation 4; CRP = C-reactive protein; dsDNA = double-stranded deoxyribonucleic acid;; FSH = follicle stimulating hormone; GGT = gamma-glutamyltransferase; HDL-C = high-density lipoprotein cholesterol; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; INR = international normalized ration; IL-21 = interleukin 21; LDL-C = low-density lipoprotein cholesterol; MAD = multiple ascending doses; MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = Mean corpuscular volume; nAb = neutralizing antibody; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; PT = prothrombin time; qual = qualitative; RBC = red blood cell; RDW = RBC distribution width; SAE = serious adverse event; SC = subcutaneous; CCI ; TB = tuberculosis.

- a On all urine samples
- At screening only, in women who are amenorrheic for at least 12 consecutive months and under 55 years old
- c For WOCBP
- d Screening only
- e At screening, and if a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium
- f Additional testing for potential Hy's Law cases only (See Section 6.2.2.6.3)
- g If patient is positive for ADA
- h If clinically indicated for hemolytic anemia

### 6.2.1.1 Pregnancy testing

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, at the last follow up visit day (Day 270) and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures (see Section 5.4) are specified in the Schedule of Assessments (see Table 1 and Table 4).

See Section 6.2.2.7.1 for information on reporting of pregnancies as AEs/SAEs during the study.

#### 6.2.1.2 Tuberculosis Screening

During the screening period, it must be determined and documented that a patient does not have evidence of active or latent or inadequately treated TB per the exclusion criteria (Section 4.5). The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the


3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).

### 6.2.1.2.1 Mycobacterium Tuberculosis Testing Using QuantiFERON Test<sup>40</sup>

QuantiFERON-TB Gold In-Tube (QFT-G) is an *in vitro* diagnostic test using a peptide cocktail simulating ESAT-6, CFP-10, and TB 7.7 proteins to stimulate cells in heparinized whole blood. Detection of INFγ performed by enzyme-linked immunosorbent assay (ELISA) is used to identify *in vitro* responses to these peptide antigens that are associated with Mycobacterium tuberculosis infection. QFT-G is an indirect test for M. tuberculosis infection (including disease) and is intended for use in conjunction with risk assessment, radiography and other medical and diagnostic evaluations.

Test results will be reported as positive, negative, or indeterminate. A negative QFT-G test result is required to meet the inclusion criterion. In the case of an indeterminate result, repeat tests should be permitted for the purpose of determining eligibility of patients to enroll in this study. If a repeat test is indeterminate again, the patient is a screen failure. The procedure for using this test and interpreting the results will be described fully in the laboratory manual, which will be provided to Investigators.

#### 6.2.2 Adverse Events

#### 6.2.2.1 Definitions

An AE is defined as any untoward medical occurrence experienced by a study patient, whether or not considered drug related by the principal Investigator.

AEs are unfavorable changes in a general condition, subjective or objective signs or symptoms, worsening of pre-existing concomitant disease, and clinically significant abnormality in laboratory parameters observed in a patient in the course of a clinical study.

Non-serious SLE manifestations or abnormal laboratory results related to SLE disease activity would not be recorded as AEs unless they meet the definition for SAEs (Section 6.2.2.5).

### 6.2.2.2 Recording of Adverse Events

AEs should be collected and recorded for each patient from the date of the first dose of study drug until the end of their participation in the study, including the safety follow up period.

AEs may be volunteered spontaneously by the study patient, or discovered by the study staff during physical examinations or by asking an open, nonleading question such as 'How have you been feeling since you were last asked?' All AEs and any required remedial action will be recorded on the Adverse Events eCRF and Safety Adverse Event Form. The details of the AE, date of AE onset, date of AE outcome, and action


taken for the AE will be documented together with the principal investigator's assessment of the seriousness of the AE and causal relationship to the study drug and/or the study procedure.

All AEs should be recorded individually, using diagnostic terms where possible. If the diagnosis is not established, individual symptoms may be reported. The AEs will subsequently be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

#### 6.2.2.3 **Severity of Adverse Events**

Each AE will be assessed by the principal Investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 criteria.41 When changes in the severity (grade) of an AE occur more frequently than once a day, the maximum severity for the event should be noted for that day. Any change in severity of signs and symptoms over a number of days will be captured by recording a new AE, with the amended severity grade and the date (and time, if known) of the change.

#### 6.2.2.4 **Causality of Adverse Events**

The principal Investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (Table 3) should be selected based on medical judgment, considering the definitions below and all contributing factors.

### **Table 3. Causality Definitions**

| Related | A clinical event, including laboratory test abnormality, occurs in a plausible time relationship to treatment administration and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (dechallenge <sup>a</sup> ) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge <sup>b</sup> procedure if necessary |
|---|---|
| Unrelated | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative dechallenge and rechallenge information. Typically explained by extraneous factors (e.g., concomitant disease, environmental factors, or other drugs or chemicals) |

- Dechallenge: Upon discontinuation of a drug suspected of causing an AE, the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation (positive dechallenge), or the symptoms continue despite withdrawal of the drug (negative dechallenge). Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia)
- Rechallenge: Upon re-administration of a drug suspected of causing an AE in a specific patient in the past, the AE recurs upon exposure (positive rechallenge), or the AE does not recur (negative rechallenge)

An unexpected adverse drug event is any adverse drug event for which the specificity or severity is not consistent with the current IP.


#### 6.2.2.5 Seriousness of Adverse Events

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life threatening; this means that the patient was at risk of death at the time of the
  event; it does not mean that the event hypothetically might have caused death if it
  were more severe
- Requires hospitalization or prolongation in existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly or birth defect
- Is other important medical event (see below)

Important medical events that do not result in death, are not life threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such events are:

- Intensive treatment in an emergency room or at home for allergic bronchospasm
- Blood dyscrasias or convulsions that do not result in inpatient hospitalization
- Development of drug dependency or drug abuse

Hospitalization for elective surgery or routine clinical procedures that are not the result of AE (e.g., elective surgery for a pre-existing condition that has not worsened) need not be considered SAEs. If anything untoward is reported during the procedure, that occurrence must be reported as an AE, either 'serious' or 'nonserious' according to the usual criteria.

Suspected unexpected serious adverse reactions (SUSARs) are AEs that are associated with the use of the drug and are serious and unexpected.

### 6.2.2.6 Adverse Events of Special Interest

AEs of special interest in this study include the following:

- 1. Anaphylaxis and serious allergic reactions
- 2. Grades 2 to 5 injection site reaction, including erythema, pain, and induration (see Appendix 6)
- 3. Drug Induced Liver Injury (DILI) assessed following Hy's Law
- 4. Malignancy (not including basal cell carcinoma or squamous cell carcinoma of skin)
- 5. Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, disseminated herpes simplex, disseminated tuberculosis, *Aspergillus* sp., *Candida albicans*, *Coccidioides immitis*, *Cryptococcus neoformans*, *Cytomegalovirus*, *Histoplasma capsulatum*, *Isospora belli*, and *Polyomavirus JC polyomavirus*


6. Cryptosporidiasis

### 6.2.2.6.1 Anaphylaxis and Serious Allergic Reactions

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria. <sup>42</sup> In the event of anaphylactic reaction or severe/serious hypersensitivity/allergic reaction, the patient must discontinue IP and emergency resuscitation measures implemented. In case of other mild to moderate hypersensitivity reaction, depending on the severity, the Investigator may manage in accordance with the standard-of-care.

Anaphylaxis is highly likely when any one of the following 3 criteria is fulfilled:

- Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (e.g., generalized hives, pruritus, or flushing, swollen lips-tongue-uvula) and at least 1 of the following:
  - a. Respiratory compromise (e.g., dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow [PEF], hypoxemia)
  - b. Reduced blood pressure or associated symptoms of end-organ dysfunction (e.g., hypotonia [collapse], syncope, incontinence)
- Two or more of the following that occur rapidly after exposure to a likely allergen for that patient (minutes to several hours):
  - a. Involvement of the skin-mucosal tissue (e.g., generalized hives, itch-flush, swollen lips-tongue-uvula)
  - b. Respiratory compromise (e.g., dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)
  - c. Reduced blood pressure or associated symptoms (e.g., hypotonia [collapse], syncope, incontinence)
  - d. Persistent gastrointestinal symptoms (e.g., crampy abdominal pain, vomiting)
- Reduced blood pressure after exposure to known allergen for that patient (minutes to several hours):
  - Systolic blood pressure of less than 90 mm Hg or greater than 30% decrease from the patient's baseline

### 6.2.2.6.2 Injection Site Reactions

Injection site reactions are to be captured and reported as AEs. These will include Grades 2 to 5 injection site erythema, pain, and induration (see Appendix 6), which are also captured as Adverse Events of Special Interest (see Section 6.2.2.6). The Investigator should provide a clear description of the observed or reported AE including location and severity. All concomitant treatments used to treat injection site reactions should be recorded and captured in the eCRF, together with the AE of injection site reactions.


#### 6.2.2.6.3 Potential Drug-Induced Liver Injury

Abnormal values in AST and/or ALT levels concurrent with abnormal elevations in total bilirubin level that meet the criteria outlined below in the absence of other causes of liver injury are considered potential cases of DILI, and as potential Hy's Law cases, and should always be considered important medical events. If symptoms compatible with DILI precede knowledge of serum chemical test abnormalities, liver enzyme measurements should be made immediately, regardless of when the next visit or monitoring interval is scheduled. In some cases, symptoms may be an early sign of injury and although typically less sensitive than serum enzyme elevations, they may indicate a need for prompt serum testing. An increase in liver enzymes should be confirmed by a repeated test within 48 to 72 hours following the initial test, prior to reporting of a potential DILI event. Patients will continue to have weekly or biweekly liver enzyme measurements until resolution or levels return to baseline.

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 6.2.2.7.2 for reporting details).

Potential DILI is defined as:

ALT or AST elevation > 3 × ULN

**AND** 

2. Total bilirubin > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)

AND

3. No other immediately apparent possible causes of ALT or AST elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic

The patient should return to the investigational site and be evaluated as soon as possible, include laboratory tests, detailed history, and physical assessment. In addition to repeating measurements of AST and ALT, laboratory tests should include albumin, CK, total bilirubin, direct and indirect bilirubin, GGT, prothrombin time (PT)/International Normalized Ratio (INR), and alkaline phosphatase. A detailed history, including relevant information, such as review of ethanol, acetaminophen, recreational drug and supplement consumption, family history, occupational exposure, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and work exposure, should be collected. Further testing for acute hepatitis A, B, or C infection and liver imaging (e.g., biliary tract) may be warranted. All cases confirmed on repeat testing as meeting the laboratory criteria defined above, with no other cause for liver function test (LFT) abnormalities identified at the time should be considered potential Hy's Law cases irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal LFTs. Such potential Hy's Law cases should be reported as SAEs.


Study drug discontinuation is considered if there is marked serum AST or ALT elevation or evidence of functional impairment (as indicated by rising bilirubin or INR, which represent substantial liver injury) that is related to study drug. Discontinuation of treatment should be considered if:

- ALT or AST > 8 × ULN
- ALT or AST > 5 × ULN for more than 2 weeks

Discontinuation of treatment must occur if:

- ALT or AST > 3 × ULN and (total bilirubin > 2 × ULN or INR > 1.5)
- ALT or AST > 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia ( > 5%)

#### 6.2.2.6.4 **Malignancy**

The identification of a malignancy event will be made by the study site and communicated to the sponsor or designee. AEs should be reported as serious per the criteria in Section 6.2.2.5.

After the first dose of study drug, when there is a decision to biopsy a potentially malignant tumor, lymph node, or other tissue (with the exception of suspected basal cell/squamous cell), the Investigator and/or consultant(s) should contact the sponsor clinicians or designee to discuss the issue and any decisions as soon as possible. Basal cell carcinoma or squamous cell carcinoma of skin is not considered an AE of special interest.

#### 6.2.2.6.5 **Specific Infections**

Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, disseminated herpes simplex, disseminated tuberculosis, Aspergillus sp., Candida albicans, Coccidioides immitis, Cryptococcus neoformans, Cytomegalovirus, Histoplasma capsulatum, Isospora belli, or Polyomavirus JC polyomavirus will be recorded as AEs of special interest.

Cryptosporidiosis is also considered an AE of special interest. Patients will be evaluated for cryptosporidium in the stool at screening, and as clinically indicated (e.g., watery diarrhea) during the study. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

#### 6.2.2.7 **Reporting of Adverse Events**

AE reporting will be carried out in accordance with applicable local regulations, including regulatory agency and IRB reporting requirements.

Each AE is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.


### 6.2.2.7.1 Reporting of Pregnancy

As information is available, a pregnancy diagnosed during the study will be reported within 24 hours to the sponsor via the Pregnancy Notification and Outcome Form, including pregnancy in female patients who received study drug and female partners of male study patients who received study drug. The pregnancy should be followed to term and/or outcome and this outcome should also be reported to the sponsor via the Pregnancy Notification and Outcome Form. Pregnancy itself is not regarded as an AE or SAE unless there is complication.

In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an AE or SAE (i.e., ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live born, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the Investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as serious adverse events when the Investigator assesses the neonatal death as related or possibly related to exposure to investigational product.

### 6.2.2.7.2 Reporting of Serious Adverse Events

The principal Investigator is responsible for providing notification to the sponsor of any SAE via the Safety Adverse Event Form, whether deemed study drug related or not, that a patient experiences during their participation in this study within 24 hours of becoming aware of the event.

If an SAE is fatal or life threatening, notification to the sponsor must be made aware immediately, irrespective of the extent of available AE information. This timeframe also applies to additional new information (follow-up) on previously forwarded SAE reports as well as to the initial and follow-up reporting of exposure during pregnancy and exposure via breastfeeding cases. In the rare event that the Investigator does not become aware of the occurrence of an SAE immediately (e.g., if an outpatient study patient initially seeks treatment elsewhere), the Investigator is to report the event within 24 hours after learning of it and document the time of his/her first awareness of the AE.

The principal Investigator will review each SAE and evaluate the intensity and the causal relationship of the event to the study drug. All SAEs will be recorded from the time of first dose of study drug through the safety follow-up period (up to Day 270).


SAEs occurring after the final follow-up visit and coming to the attention of the principal Investigator must be reported only if there is (in the opinion of the principal Investigator)

reasonable causal relationship with the study drug.

As a minimum requirement, the initial notification should provide the following information:

Study number

- Patient number
- Details of the SAE (verbatim details are sufficient for immediate notification)
- Criterion for classification as 'serious'
- Causality assessment (which may be updated in a follow-up report when sufficient information is available to make this classification)

Initial reports of SAEs must be followed later with detailed descriptions, including clear photocopies of other documents as necessary (e.g., hospital reports, consultant reports, autopsy reports, etc), with the study patient's personal identifiers removed. All relevant information obtained by the principal Investigator through review of these documents will be recorded and submitted to the sponsor within 24 hours of receipt of the information. If a new Safety Adverse Event Form is submitted, then the principal Investigator must sign and date the form. The sponsor may also request additional information on the SAE, or clarification of omitted or discrepant information from the initial notification, which the principal Investigator or an authorized delegate should submit to the sponsor within 24 hours of the request as possible.

### 6.2.2.7.3 Reporting of Adverse Events of Special Interest

AEs of special interest will be reported to safety immediately or within 24 hours of the site becoming aware of the event and recorded as such on the Adverse Events eCRF and Safety Adverse Event Form.

Potential DILI will be reported based on specifications mentioned in Section 6.2.2.6.3.

Each AE of special interest is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

### 6.2.2.8 Follow Up of Adverse Events

All AEs will be followed up through the safety follow-up visits. All SAEs experienced by a patient, irrespective of the suspected causality, will be monitored until the event has resolved, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the principal Investigator and medical monitor, until there is a satisfactory explanation for the changes observed, or until the patient is lost to follow-up.


See Section 6.2.2.7.1 for details related to follow-up of pregnancy. See Section 6.2.2.6.3 for details related to follow-up of potential DILI. See Section 6.2.2.6.4

for details related to follow-up of malignancy.

### 6.2.3 Vital Signs

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (Table 1 and Table 4). Vital signs will be assessed on Day 0 at predose and at Day 0, 1 and 2 hours ( $\pm$  15 minutes) postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq$  5 minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

### 6.2.4 12-Lead Electrocardiograms

ECG will be assessed as specified in the Schedule of Assessments (Table 1 and Table 4). ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

The ECG will include all 12 standard leads and a Lead II rhythm strip on the bottom of the tracing. The ECG will be recorded at a paper speed of 25 mm/second. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QT interval corrected for heart rate using Fridericia's formula (QTcF).

All ECGs must be evaluated by a qualified physician or qualified designee for the presence of abnormalities and will be captured electronically and retained for future evaluation if required, up to the time of the clinical study report (CSR) completion.

#### 6.2.5 Physical Examinations

The full physical examination will be completed at screening and Day 0. It includes an assessment of general appearance and evaluation of head, eyes, ears, nose, mouth, throat, neck, thyroid, lymph nodes, and extremities, and dermatologic, respiratory, cardiovascular, gastrointestinal, musculoskeletal, neurologic, and psychiatric systems.

The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Table 1 and Table 4). It includes evaluation of patient complaints and SLE disease-related issues, and will exclude the genitourinary system.

#### 6.2.6 C-SSRS

The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed by Columbia University researchers for the National Institute of


Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening.<sup>43</sup>

The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Table 1 andTable 4). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

### 6.2.7 Injection Site Reactions

Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (Table 1 and Table 4). Local injection site reactions will be assessed at 2 hours postdose at baseline, and predose for each injection after baseline. Injection site reactions should be managed according to the standard of care. Injection site reactions, Grades 2 to 5, are to be reported as AEs of special interest (see Section 6.2.2.7.3).

### 6.2.8 Immunogenicity

The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (Table 1 and Table 4). Blood samples (4 mL) to provide approximately 1.5 mL of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K<sub>2</sub>EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only analyzed by a central lab if the patient had a positive ADA on Day 90.

After the first dose, if a patient tests positive in the validated confirmatory ADA assay, a sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay by a central lab.

### **6.3 Efficacy Assessments**

All efficacy assessments will be performed at times defined in the Schedule of Assessments (Table 1 and Table 4).

#### 6.3.1 SLEDAI-2K

The SLEDAI-2K is a validated instrument that measures disease activity in SLE patients at the time of the visit and in the previous 30 days. It is a global index and includes 24 clinical and laboratory variables that are weighted by the type of manifestation, but


not by severity. The total score falls between 0 and 105, with higher scores representing increased disease activity. The SLEDAI-2K has been shown to be a valid and reliable disease activity measure in multiple patient groups. A SLEDAI -2K of 6 or more generally represents moderately to severely active disease.<sup>44</sup>

#### 6.3.2 BILAG 2004

The BILAG-2004 index is an organ-specific 97-question assessment based on the principle of the doctor's intent to treat. Only clinical features attributable to SLE disease activity are to be recorded and based on the patient's condition in the last 4 weeks compared with the previous 4 weeks. It will be scored as not present (0), improved (1), the same (2), worse (3), or new (4). Disease activity is graded separately for 9 body systems to 5 different grades (A to E) as follows: A ("Active") is very active disease, B ("Beware") is moderate activity, C ("Contentment") is mild stable disease, D ("Discount") is inactive now but previously active, and E ("Excluded") indicates the organ was never involved. A shift from BILAG-2004 Grade A or B to a lower grade indicates a clinically relevant change in disease activity as the BILAG-2004 grades mirror the decision points for treatment interventions.

Only Investigators that complete BILAG-2004 training will be allowed to perform the BILAG-2004 assessments. Preferably, the same Investigator should evaluate the patient at each BILAG-2004 assessment from screening to study completion. The Investigator must maintain documentation with descriptive details supporting the BILAG-2004 scoring (e.g., chart, worksheet, clinic notes, and labs) at each visit.

See Appendix 5 for detailed specifications.

#### 6.3.3 PGA of Disease Activity

The PGA is used to assess Investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients". PGA worsening is defined as an increase of > 30 mm from baseline.

When scoring the PGA, the assessor should always look back at the score from the previous visit.

#### 6.3.4 Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response

#### 6.3.4.1 SRI-4 Response

The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. Response based on the SRI-4 is defined by:

1)  $\geq$  4-point reduction in SLEDAI-2K global score; 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B); and 3) no


deterioration from baseline in the PGA by  $\geq$  30 mm. The SRI-4 response in patients with moderate to severe SLE is associated with broad improvements in clinical and patient-reported outcomes.<sup>45</sup>

### 6.3.4.2 SRI-5 and SRI-6 Response

Like the SRI-4, the SRI-5 and SRI-6 are composite indices of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. However, the SRI-5 and SRI-6 are computed with a minimal five-point or six-point improvement in SLEDAI-2K being required, respectively.<sup>46</sup>

### 6.3.4.3 BICLA Response

The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and PGA. BICLA response is defined as: 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (e.g., all B [moderate disease] scores falling to C [mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4)  $\leq$  10% deterioration in PGA score; and 5) no treatment failure.<sup>44</sup> It is driven primarily by the BILAG, and has been used in phase 2 and 3 mAb studies.<sup>47</sup>

For the endpoints of BICLA response at Days 210, 240, and 270, patient scores will be completed and response determined.

#### 6.3.5 CLASI Response

The CLASI is a comprehensive tool for assessment of disease activity and damage in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity.<sup>48</sup> Response is defined as 50% improvement from baseline in "A" or "B" scores. This assessment will be applied to all patients who have cutaneous disease activity.

For the secondary efficacy endpoint of CLASI response at Day 210, patient scores on MAD and POC studies will be compared with baseline for 50% improvement.

### 6.3.6 ACR-28 Joint Count

The ACR-28 joint count will evaluate the number of tender and swollen joints in the shoulder, elbow, wrist, hand, knee joints. Joints of the feet are excluded.

#### 6.4 Other Variables

#### 6.4.1 SLICC/ACR Damage Index

The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in patients with SLE regardless of cause,


with demonstrated content, face, criterion, and discriminant validity.<sup>49</sup> It will be performed on Days 0 and 180.

#### 6.4.2 PROs

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the and the and will be assessed as specified in the Schedule of Assessments (Table 1 and Table 4).



#### 6.5 Pharmacokinetic Assessments

During the MAD phase 1b (all sites) and POC phase 2 (select sites only) parts of the study, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to Table 4 and Table 1.

Plasma concentrations of BOS161721 will be measured using a validated immunoassay. The PK parameters will be calculated from the plasma concentration actual time profiles.

### 6.6 Pharmacodynamic Assessments

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (Table 1 and Table 4) for each of the following parameters:

- pSTAT3 (predose [trough] samples only phase 1b)
- Antibodies: CCI
- Plasma complement (CCI)
- Plasma CCI and CCI
- Whole blood for leukocyte immunophenotype (for MAD patients only)

# 6.7 Pharmacokinetic/Pharmacodynamic Relationship

Evidence of any PK/PD relationships will be evaluated between BOS161721 plasma concentrations and the available PD endpoints and biomarkers.


#### 6.8 Protocol Deviations

Protocol deviations will be documented during the study.

#### 7 STUDY DRUG MANAGEMENT

### 7.1 Description

#### 7.1.1 Formulation



Additional information regarding dose preparation will be provided in a separate Pharmacy Manual.

#### 7.1.2 Storage

All supplies of BOS161721 or placebo must be stored in accordance with the manufacturer's instructions. BOS161721 or placebo will be stored in a securely locked area, accessible to authorized persons only, until needed for dosing.

Information regarding storage and dose preparation will be provided in a separate Pharmacy Manual.

### 7.2 Packaging and Shipment

Investigational medicinal products will be supplied by Boston Pharmaceuticals, Inc. Investigational medicinal products will be packaged and labeled according to applicable local and regulatory requirements.

#### 7.3 Dose and Administration

receive the matching number of kits.

Details of dosing are provided in Section 3.1.

Each unit dose will be prepared by a qualified staff member. The vials of investigational product (IP) will appear identical and will have a "blinded" label on the vials that will state mg or placebo. When the site goes into the IWRS to request the patient kit(s), the IWRS will assign the appropriate number of kits (regardless of assignment to placebo or active treatment) per the dose (i.e., CCI). If a patient is randomized to the placebo arm, they will


The designated staff member (or designee under the direction of the designated staff member) will dispense BOS161721 or placebo for each patient according to the protocol, randomization list, and Pharmacy Manual, if applicable.

After receiving sponsor approval in writing, the investigational site is responsible for returning all unused or partially used BOS161721 or placebo to the sponsor or designated third party or for preparing BOS161721 or placebo for destruction via incineration.

Further details are found in a separate Pharmacy Manual.

### 7.4 Accountability

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed, and amount returned to the pharmacy (if any). Used investigational product returned to the pharmacy may be maintained in an ambient condition. Unused product should follow the instructions in the Pharmacy Manual. The used product that is returned should be marked as 'returned' and kept separate from the products not yet dispensed.

All dispensing and accountability records will be available for sponsor review after database lock procedures are completed. During safety monitoring, the drug accountability log will be reconciled with the products stored in the pharmacy.

### 7.5 Prohibited Concomitant Therapy

Prohibited concomitant medications are discussed in Section 4.6 and Appendix 4 will be listed as protocol violations if taken when not permitted.

## 7.6 Compliance

Dosing will be performed by trained, qualified personnel designated by the principal Investigator. The date and time of dosing will be documented on each dosing day. Comments will be recorded if there are any deviations from the planned dosing procedures.

#### 8 STATISTICS

The following analyses are planned:

- An IA will be performed during the last cohort of the MAD portion to determine dose selection for the POC part of the study.
- An additional analysis may be performed for the MAD portion of the study when all MAD patients have completed the safety follow-up or withdrawn from the study, and


prior to final analysis. Data from the POC part of the study will be excluded from this additional analysis.

- The final analysis will be performed when all patients have completed the POC safety follow-up or withdrawn from the study.
- Safety analyses will be performed for DMC reviews throughout the study to evaluate dose escalation decisions and accumulating safety data. The frequency and details of the content and format of the safety review meetings will be described in the SAP and/or DMC charter.

All statistical analyses will be performed using Statistical Analysis Software (SAS®) Version 9 or higher.

The following standards will be applied for the analysis unless otherwise specified. Data will be summarized descriptively by treatment and overall for each study portion. For the MAD part of the study, BOS161721 will be summarized overall and by each dose level, and placebo patients from each cohort will be combined. Select parameters may be summarized using patients from both study parts. Statistical testing will be performed on data from the phase 2 portion only.

Continuous data will be summarized using number, mean, standard deviation (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, median, and maximum. Categorical data will be summarized by treatment group using frequency tables (number and percentage). Time to event data will be summarized using counts, medians, 25<sup>th</sup> and 75<sup>th</sup> percentiles, and standard error. All data will be listed for all patients.

Statistical inference will be based on a 2-tailed test with an overall 0.10 level of significance, unless stated otherwise.

The effects of noncompliance, background therapy use, treatment discontinuations, premature withdrawal from study and covariates will be assessed to determine the impact on the general applicability of results from this study. Exploratory analyses of the data will be conducted as deemed appropriate. Any deviations from the planned analyses will be described and justified in the final integrated CSR.

Protocol deviations and prohibited medications that define medication failures will be fully assigned and documented before database lock and unblinding.

Further details of the analysis, including the handling of missing data, transformations and other data handling procedures will be provided in the SAP.

### 8.1 Sample Size

Sample size in the phase 1b part of the study is based on operational consideration.

The sample size in the phase 2 portion is based on the primary endpoint, SRI-4 Response at Day 210. Based on efficacy data from a recently completed study with Ustekinumab<sup>51</sup>, where the primary endpoint was also SRI-4, the sample size in the phase 2 part of the BOS161721-02 study is set at 96 evaluable patients. In the


Ustekinumab study of 102 patients, a statistically significant difference in SRI-4 response was shown in favor of Ustekinumab (62% of Ustekinumab treated patients achieved SRI-4 response vs. 33% in patients receiving placebo). The Ustekinumab phase 2 study is an appropriate comparator to BOS161721-02 because both studies share the same primary endpoint of SRI-4 response and BOS161721 and Ustekinumab have overlapping mechanisms of action (T follicular helper and Th17 cell biology).

Approximately 110 additional patients will be randomized in a 2:1 ratio to BOS161721 versus placebo to achieve approximately 96 evaluable patients in the FAS of the phase 2 portion. This assumes 14 patients will drop prior to having received treatment or having completed a post-baseline efficacy measure. Enrollment and randomization will be monitored in a blinded fashion and may be increased if needed to ensure at least 96 evaluable patients are randomized into the FAS.

A total of 96 evaluable patients randomized provides 80% power to detect a treatment difference of 29% in SRI-4 response rates at Day 210, based on a targeted 2-sided significance level of 10% and using a 2-sided Pearson's chi-squared test. This assumes a response rate of 62% for BOS161721 and 33% for placebo.

#### 8.2 Statistical Methods

### 8.2.1 Analysis Populations

The primary efficacy analysis will be based on the FAS, defined as all patients who receive at least 1 dose (partial or complete) of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. FAS analyses will be conducted on the basis of the randomized treatment.

A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be identified based on blinded data prior to study unblinding. PP analyses will be conducted on the basis of the randomized treatment.

Safety analyses will be based on the safety analysis set (SS), defined as all patients who receive at least 1 dose (partial or complete) of study treatment. Safety analyses will be conducted on the basis of actual treatment received.

Pharmacokinetic analysis will be conducted on the PK analysis set, defined as the FAS with sufficient concentration data for the calculation of PK parameters.

#### 8.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized using all randomized patients.


### 8.2.3 Primary Efficacy Endpoint(s)

The proportion of patients who achieve a SRI-4 response at Day 210 will be assessed via Pearson's chi-squared analysis. The primary efficacy endpoint will be analyzed using the FAS and if needed repeated in the PP analysis set. Missing values will be addressed by employing a last observation carried forward (LOCF) analysis. Other imputation methods may be employed as a sensitivity analysis and will be described in the SAP. Analyses based on observed values may also be performed.

Exploratory subgroup analyses assessing impact of baseline factors such as baseline disease severity, background therapy, race, geography, baseline serologic activity and other characteristics may be performed. Additional exploratory analyses of disease activity endpoints may be performed based on emerging data.

Patients that received prohibited medications or unallowable CS usage as described in Section 4.6 will be considered "medication failures" and will be treated as statistical non-responders at time points on or following the first date of prohibited medication or unallowable CS usage for the primary efficacy analysis. The determination of medication failures will be reviewed using blinded data and finalized prior to unblinding.

The superiority of BOS161721 relative to placebo will be evaluated. If the proportion of SRI-4 responders for the selected POC dose in BOS161721 arm is higher than that of the placebo arm, then BOS161721 will be considered superior to placebo if the 2-sided p-value is < 0.10. Secondary and exploratory endpoints for this POC portion will be evaluated based on the same statistical hypothesis.

#### 8.2.4 Secondary Efficacy Endpoint(s)

Binary efficacy endpoints will be assessed via Pearson's chi-squared analysis. Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) and treatment will be compared using the F-test. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test. The secondary efficacy endpoints will be analyzed on the FAS and if needed repeated in the PP analysis set. Details including handling of missing data and "medication failures" will be available in the SAP.

### 8.2.5 Analysis of Safety

#### 8.2.5.1 Safety Analysis

Safety analyses will be performed on the SS. AE data will be coded to system organ class and preferred term using MedDRA. The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term, will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.


Concomitant medications will be coded using the WHO Drug dictionary. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters will be summarized at each individual visit.

### 8.2.6 Pharmacokinetic and Pharmacodynamic Data

### 8.2.6.1 Analysis of Pharmacokinetic Data

PK parameters will be calculated from concentration data collected during the MAD phase 1b portion of the study using non-compartmental analysis and include the following:

• C<sub>max</sub>, T<sub>max</sub>, AUC, t<sub>1/2</sub>, CL, V<sub>d</sub>

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:

- A listing of all plasma BOS161721 concentrations by patient at actual times post dose;
- A descriptive summary of plasma BOS161721 concentrations. Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.

### 8.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Exploratory analyses examining the relationship between PD parameters and PK concentration and PK parameters will be performed.

### 8.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints.

## 8.3 Interim Analysis and Power

One IA is planned for this study and will be conducted at the time of the POC decision for dose selection.

Since there is no IA during the POC part of the study, there is no impact on the type 1 error.


#### 9 ETHICS AND RESPONSIBILITIES

#### 9.1 Good Clinical Practice

The procedures set out in this protocol are designed to ensure that the sponsor and the principal Investigator abide by the principles of the International Council for Harmonisation (ICH) guidelines on GCP and the Declaration of Helsinki (Version 2013). The clinical study also will be carried out in the keeping with national and local legal requirements (in accordance with US IND regulations [21 CFR 56]).

#### 9.2 DMC

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for BOS161721. The recommendations made by the DMC (i.e., dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.

The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study Investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) suggest dose for POC portion of the study as described in Section 3.1.1.3.

The DMC considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

The DMC will have access to unblinded treatment information during the clinical trial. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of BOS161721 treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential


benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.

### 9.3 Institutional Review Board/Independent Ethics Committee

Independent Ethics Committees/IRB must meet the guidelines set out by the U. S. Food and Drug Administration (FDA) and conform to local laws and customs where appropriate. Written IRB/IEC approval for the protocol and the signed ICF must be obtained and transmitted to Boston Pharmaceuticals or representative before the study can be initiated. The IRB/IEC must be informed of and approve all protocol amendments. The Investigator will ensure that this study is conducted in full conformance with all applicable local and regional laws and regulations. The complete text of the World Medical Association Declaration of Helsinki is given in Appendix 2.

#### 9.4 Informed Consent

Before each patient undergoes any protocol required assessments or procedure, the written informed consent will be obtained according to the regulatory and legal requirements of the participating country. As part of this procedure, the principal Investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study patient should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The principal Investigator or designee will provide the sponsor with a copy of the IRB-approved ICF prior to the start of the study.

The informed consent document must be signed and dated; 1 copy will be handed to the patient and the principal Investigator will retain a copy as part of the clinical study records. The principal Investigator will not undertake any investigation specifically required for the clinical study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented.

If the informed consent document is revised, it must be reviewed and approved by the responsible IRB/IEC. Patients currently enrolled may need to sign this revision (based on IRB/IEC requirements) and all future patients enrolled in the clinical study will be required to sign this revised ICF.

### 9.5 Records Management

The principal Investigator will ensure the accuracy, completeness, and timeliness of the data reported to the sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes. The principal Investigator or designee will cooperate with the sponsor's representative(s) for the periodic review of study documents to ensure the accuracy and completeness of the data capture system at each scheduled monitoring visit.


Electronic consistency checks and manual review will be used to identify any errors or inconsistencies in the data. This information will be provided to the respective study sites by means of electronic or manual queries.

The principal Investigator or designee will prepare and maintain adequate and accurate study documents (medical records, ECGs, AE and concomitant medication reporting, raw data collection forms, etc.) designed to record all observations and other pertinent data for each patient receiving BOS161721 or placebo.

The principal Investigator will allow sponsor representatives, contract designees, authorized regulatory authority inspectors, and the IRB to have direct access to all documents pertaining to the study.

Electronic case report forms are required and should be completed for each randomized patient. It is the principal Investigator's responsibility to ensure the accuracy, completeness, legibility, and timeliness of the data reported on the patients' eCRF. Electronic case report forms should be completed in a timely fashion to support the study timelines. Source documentation supporting the eCRF data should indicate the patient's participation in the study and should document the dates and details of study procedures, AEs, and patient status. The principal Investigator or designated representative should complete and the principal Investigator should verify the source documents as the information is collected. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

The principal Investigator will ensure the accuracy, completeness, and timeliness of the data reported to the Sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes.

#### 9.6 Source Documentation

The documents that will form the source data for the clinical study (e.g., patient charts, laboratory reports) must be defined and documented in the in-house study master file prior to the start of the study. Data on the eCRFs which will be checked against source data during monitoring visits must also be defined and documented in the in-house study master file including the percentage of each of the source data to be verified and the percentage of patients' eCRFs to be monitored.

# 9.7 Study Files and Record Retention

According to ICH guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of BOS161721. However, these documents should be retained for a longer period if required by the applicable legal requirements.


#### 10 AUDITING AND MONITORING

Throughout the course of the study, the study monitor will make frequent contacts with the Investigator. This will include telephone calls and on-site visits. The study will be routinely monitored to ensure compliance with the study protocol and the overall quality of data collected. During the on-site visits, the eCRFs will be reviewed for completeness and adherence to the protocol. As part of the data audit, source documents will be made available for review by the study monitor. The study monitor may periodically request review of the Investigator study file to assure the completeness of documentation in all respects of clinical study conduct. The study monitor will verify that each patient has proper consent documentation from the patient and/or patient's authorized representative for study procedures and for the release of medical records to the sponsor, FDA, other regulatory authorities, and the IRB. The study monitor will also verify that assent was obtained for patients not capable of providing informed consent or that documentation is provided by the Investigator explaining why the patient was unable to provide assent. The Investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the Investigator will permit inspection of the study files by authorized representatives of the regulatory agencies. On completion of the study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

Throughout the course of the study, the medical monitor will determine eligibility of all screened patients, will address any medical issues that might arise, clarify medical questions, review patient safety data (e.g., AE/SAE, laboratory, and ECG), and partner with the study team in the overall study management. The study medical monitoring plan will document additional details of the study medical oversight and monitoring.

#### 11 AMENDMENTS

Protocol modifications, except those intended to reduce immediate risk to study patients, may be made only by Boston Pharmaceuticals. A protocol change intended to eliminate an apparent immediate hazard to patients may be implemented immediately, provided the IRB/IEC is notified within 5 days.

Any permanent change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB/IEC and the Investigator must await approval before implementing the changes. Boston Pharmaceuticals will submit protocol amendments to the appropriate regulatory authorities for approval.

If in the judgment of the IRB/IEC, the Investigator, and/or Boston Pharmaceuticals, the amendment to the protocol substantially changes the study design and/or increases the potential risk to the patient and/or has an impact on the patient's involvement as a study participant, the currently approved written ICF will require similar modification. In such cases, informed consent will be renewed for patients enrolled in the study before continued participation.


#### 12 STUDY REPORT AND PUBLICATIONS

Boston Pharmaceuticals is responsible for preparing and providing the appropriate regulatory authorities with clinical study reports according to the applicable regulatory requirements.

By signing the protocol, the principal Investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the principal Investigator's name, address, qualifications, and extent of involvement.

The principal Investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted and obtained approval from the sponsor in advance.

#### 13 STUDY DISCONTINUATION

Both Boston Pharmaceuticals and the principal Investigator reserve the right to terminate the study at the Investigator's site at any time. Should this be necessary, Boston Pharmaceuticals or a specified designee will inform the appropriate regulatory authorities of the termination of the study and the reasons for its termination, and the principal Investigator will inform the IRB/IEC of the same. In terminating the study Boston Pharmaceuticals and the principal Investigator will assure that adequate consideration is given to the protection of the patients' interests.

#### 14 CONFIDENTIALITY

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from Boston Pharmaceuticals, except to the extent necessary to obtain informed consent from patients who wish to participate in the trial or to comply with regulatory requirements. However, authorized regulatory officials, IRB/IEC personnel, Boston Pharmaceuticals, and its authorized representatives are allowed full access to the records.

Identification of patients and eCRFs shall be by initials, birthdate, or patient number. Documents that identify the patient (e.g., the signed informed consent document) must be maintained in confidence by the principal Investigator. If required, the patient's full name may be made known to an authorized regulatory agency or other authorized official.


#### 15 REFERENCES

- 1 Urowitz MB, Gladman DD. How to improve morbidity and mortality in systemic lupus erythematosus. Rheumatology 2000;39:238-44.
- 2 Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, et al. Morbidity and Mortality in Systemic Lupus Erythematosus During a 10-Year Period. Medicine 2003;82(5):299-308.
- 3 Pons-Estel GJ, Alarcón GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010;39(4):257. Epub 2009 Jan 10.
- 4 Kanta H, Mohan C. Three Checkpoints in lupus development: central tolerance in adaptive immunity, peripheral amplification by innate immunity, and end-organ inflammation. Genes and Immunity 2009;10:390-6.
- 5 Dall'Aqua WF, Kiener PA, Wu H. Properties of Human IgG1s Engineered for Enhanced Binding to the Neonatal Fc Receptor (FcRn). J Biol Chem. 2006 Aug 18, 281(33):23514-24.
- 6 Spolski R, Leonard WJ. The Yin and Yang of interleukin-21 in allergy, autoimmunity and cancer. Curr Opin Immunol. 2008a;20:295-301.
- 7 Asao H, Okuyama C, Kumaki S, Ishii N, Tsuchiya S, Foster D, et al. Cutting edge: the common gamma-chain is an indispensable subunit of the IL-21 receptor complex. J Immunol. 2001;167:1-5.
- 8 Habib T, Senadheera S, Weinberg K, Kaushansky K. The common gamma chain (gamma c) is a required signaling component of the IL-21 receptor and supports IL-21-induced cell proliferation via JAK3. Biochemistry. 2002;41:8725-31.
- 9 Spolski R, Leonard WJ. Interleukin-21: basic biology and implications for cancer and autoimmunity. Annu Rev Immunol. 2008b;26:57-79.
- 10 Puga I, Cols M, Barra CM, He B, Cassis L, Gentile M, et al. B-cell-helper neutrophils stimulate the diversification and production of immunoglobulin in the marginal zone of the spleen. Nat Immunol. 2011;13(2):170-80.
- 11 Costanzo A, Chimenti MS, Botti E, Caruso R, Sarra M, Monteleone G. IL-21 in the pathogenesis and treatment of skin diseases. J Dermatol Sci. 2010;60(2):61-6.
- 12 Avery DT, Bryant VL, Ma CS, de Waal Malefy R, Tangye SG. IL-21-induced isotype switching to IgG and IgA by human naive B cells is differentially regulated by IL-4. J Immunol. 2008;181:1767-79.
- 13 Rasmussen TK, Andersen T, Bak, RO, Yiu G, Sorensen CM, Stengaard-Pedersen K, et al. Overexpression of microRNA-155 increases IL-21 mediated STAT3 signaling and IL-21 production in systemic lupus erythematosus. Arthritis Research & Therapy 2015;17(154)


- 14 Ettinger R, Kuchen S, Lipsky PE. The role of IL-21 in regulating B-cell function in health and disease. Immunol Rev. 2008;223:60-86.
- 15 Caprioli F, Sarra M, Caruso R, Stolfi C, Fina D, Sica G, et al. Autocrine regulation of IL-21 production in human T lymphocytes. J Immunol. 2008;180(3):1800-7.
- 16 Yang L, Anderson DE, Baecher-Allan C, Hastings WD, Bettelli E, Oukka M, et al. IL-21 and TGF-beta are required for differentiation of human T(H)17 cells. Nature. 2008;454(7202):350-2.
- 17 Tangye SG, Ma CS, Brink R, Deenick EK. The good, the bad and the ugly TFH cells in human health and disease. Nat Rev Immunol. 2013;13(6):412-26.
- 18 Fantini MC, Rizzo A, Fina D, Caruso R, Becker C, Neurath MF, et al. IL-21 regulates experimental colitis by modulating the balance between Treg and Th17 cells. Eur J Immunol. 2007;37(11):3155-63.
- 19 Peluso I, Fantini MC, Fina D, Caruso R, Boirivant M, MacDonald TT, et al. IL-21 counteracts the regulatory T-cell-mediated suppression of human CD4+ T lymphocytes. J Immunol. 2007;178(2):732-9.
- 20 Hippen KL, Bucher C, Schirm DK, Bearl AM, Brender T, Mink KA, et al. Blocking IL-21 signaling ameliorates xenogeneic GVHD induced by human lymphocytes. Blood. 2012;119(2):619-28.
- 21 Davis ID, Skrumsager BK, Cebon J, Nicholaou T, Barlow JW, Moller NP, et al. An open- label, two-arm, phase I trial of recombinant human interleukin-21 in patients with metastatic melanoma. Clin Cancer Res. 2007;13:3630-6.
- 22 Frederiksen KS, Lundsgaard D, Freeman JA, Hughes SD, Holm TL, Skrumsager BK, et al. IL-21 induces in vivo immune activation of NK cells and CD8(+) T-cells in patients with metastatic melanoma and renal cell carcinoma. Cancer Immunol Immunother. 2008;57(10):1439-49.
- 23 Karrich JJ, Jachimowski LC, Nagasawa M, Kamp A, Balzarolo M, Wolkers MC, et al. IL-21- stimulated human plasmacytoid dendritic cells secrete granzyme B, which impairs their capacity to induce T-cell proliferation. Blood. 2013;121(16):3103-11.
- 24 Lindner S, Dahlke K, Sontheimer K, Hagn M, Kaltenmeier C, Barth TF, et al. Interleukin-21-induced granzyme B-expressing B-cells infiltrate tumors and regulate T-cells. Cancer Res. 2013;73(8):2468-79.
- 25 Monteleone G, Caruso R, Fina D, Peluso I, Gioia V, Stolfi C, et al. Control of matrix metalloproteinase production in human intestinal fibroblasts by interleukin 21. Gut. 2006;55(12):1774-80.
- 26 Nakou M, Papadimitraki ED, Fanouriakis A, Bertsias GK, Choulaki C, Goulidaki N, et al. Interleukin-21 is increased in active systemic lupus erythematosus patients and contributes to the generation of plasma B-cells. Clin Exp Rheumatol. 2013;31(2):172-9.


- 27 Li Q, Liu Z, Dang E, Jin L, He Z, Yang L, et al. Follicular helper T-cells (Tfh) and IL-21 involvement in the pathogenesis of bullous pemphigoid. PLoS One. 2013;8(7):e68145.
- 28 Liu R, Wu Q, Su D, Che N, Chen H, Geng L, et al. A regulatory effect of IL-21 on T follicular helper-like cell and B-cell in rheumatoid arthritis. Arthritis Res Ther. 2012;14(6):R255.
- 29 Kang KY, Kim HO, Kwok SK, Ju JH, Park KS, Sun DI, et al. Impact of interleukin-21 in the pathogenesis of primary Sjögren's syndrome: increased serum levels of interleukin-21 and its expression in the labial salivary glands. Arthritis Res Ther. 2011;13(5):R179.
- 30 Terrier B, Geri G, Chaara W, Allenbach Y, Rosenzwajg M, Costedoat-Chalumeau N, et al. Interleukin-21 modulates Th1 and Th17 responses in gianT-cell arteritis. Arthritis Rheum. 2012a;64(6):2001-11.
- 31 Terrier B, Costedoat-Chalumeau N, Garrido M, Geri G, Rosenzwajg M, Musset L, et al. Interleukin 21 correlates with T-cell and B-cell subset alterations in systemic lupus erythematosus. J Rheumatol. 2012b;39(9):1819-28.
- 32 International Conference on Harmonisation. Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals S6 (R1). 2011.
- 33 Wang W, Wang EQ, Balthasar JP. Monoclonal Antibody Pharmacokinetics and Pharmacodynamics. Clin Pharm & Ther 2008; 84(5):548-58.
- 34 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 35 Elsaesser H, Sauer K, Brooks DG. IL-21 is required to control chronic viral infection. Science. 2009;324(5934):1569-72.
- 36 Kotlarz D, Zietara N, Uzel G, Weidemann T, Braun CJ, Diestelhorst J, et al. Loss-of-function mutations in the IL-21 receptor gene cause a primary immunodeficiency syndrome. J Exp Med. 2013;210(3):433-43.
- 37 Hunter PR, Nichols G. Epidemiology and clinical features of Cryptosporidium infection in immunocompromised patients. Clinical microbiology reviews. 2002;15(1):145-54.
- 38 Desjardins M, Mazer BD. B-cell memory and primary immune deficiencies: interleukin-21 related defects. Curr Opin Allergy Clin Immunol. 2013;13(6):639-45.
- 39 Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron.1976;16(1):31-41.


40 Guidelines for Using the QuantiFERON®-TB Gold Test for Detecting Mycobacterium tuberculosis Infection, US: http://www. cdc. gov/mmwr/preview/mmwrhtml/rr5415a4. htm.

- 41 NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, available at https://evs. nci. nih. gov/ftp1/CTCAE/About. html.
- 42 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 43 Posner K, Melvin G a, Stanley B, Oquendo M a, Gould M. Factors in the assessment of suicidality in youth. CNS Spectr. 2007;12(2):156-162.
- 44 Castrejon I, Tani C, Jolly M, Huang A, Mosca M. Indices to assess patients with systemic lupus erythematosus in clinical trials, long-term observational studies, and clinical care. Clin Exp Rheumatol 2014; 32(85):S85-95.
- 45 Furie R, Wang L, Drappa J, Illei G. Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] Response Is Associated with Global Benefit in Patients with Moderate to Severe SLE [abstract]. Arthritis Rheumatol. 2016; 68 (suppl 10).
- 46 Thanou A, Chakravarty E, James JA, Merrill JT. Which outcome measures in SLE clinical trials best reflect medical judgment? Lupus Science & Medicine 2014;1:e000005. doi:10.1136/lupus-2013-000005.
- 47 Wallace DJ, Kalunian K, Petri MA, Strand V, Houssiau FA, Pike M,et al. Efficacy and safety of epratuzumab in patients with moderate/severe active systemic lupus erythematosus: results from EMBLEM, a phase IIb, randomised, double-blind, placebo-controlled, multicentre study. Ann Rheum Dis 2014;73:183-90.
- 48 Albrecht J, Taylor L, Berlin JA, Dulay S, Ang G, Fakharzadeh S. The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index): An Outcome Instrument for Cutaneous Lupus Erythematosus. J Invest Derm. 2005;125(5):889-94.
- 49 Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is Valid, and Renal and Pulmonary Organ Scores are Predictors of Sever Outcome in Patients with Systemic Lupus Erythematosus. Br J Rheumatol.1996;35:248-54.

50 CCI

51 Van Vollenhoven RF, Hahn BH, Tsokos GC, et al. Efficacy and safety of ustekinumab, an IL-12 and IL-23 inhibitor, in patients with active systemic lupus erythematosus: results of a multicentre, double-blind, phase 2, randomised, controlled study. Lancet. 2018;392(10155):1330-1339.


BOS161721 Boston Pharmaceuticals, Inc


# **16 APPENDICES**


### 16.1 Appendix 1: Names of Study Personnel




### 16.2 Appendix 2: Declaration of Helsinki

#### WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI

Ethical Principles For Medical Research Involving Human Subjects.

Adopted by the 18th WMA General Assembly
Helsinki, Finland, June 1964
and amended by the
29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
and the
52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### A. INTRODUCTION

The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.

It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.

The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my subject will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the subject's interest when providing medical care which might have the effect of weakening the physical and mental condition of the subject".

Medical progress is based on research, which ultimately must rest in part on experimentation involving human subjects.

In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.

The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic, and therapeutic procedures and the understanding of the etiology and pathogenesis of disease. Even the best-proven prophylactic, diagnostic, and therapeutic methods must continuously be challenged through research for their effectiveness, efficiency, accessibility, and quality.

In current medical practice and in medical research, most prophylactic, diagnostic, and therapeutic procedures involve risks and burdens.


Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.

Research Investigators should be aware of the ethical, legal, and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal, or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### B. BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.

Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.

Appropriate caution must be exercised in the conduct of research, which may affect the environment, and the welfare of animals used for research must be respected.

The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the Investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any SAEs. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.

The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles enunciated in this Declaration.

Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a subject of the research, even though the subject has given consent.


Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.

Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.

Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.

Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.

The subjects must be volunteers and informed participants in the research project.

The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the subject's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.

In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.

When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.

For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the Investigator must obtain informed consent from the legally authorized representative in accordance with applicable law. These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.


When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the Investigator must obtain that assent in addition to the consent of the legally authorized representative.

Research on individuals from whom it is not possible to obtain consent, including proxy or advance consent, should be done only if the physical/mental condition that prevents obtaining informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.

Both authors and publishers have ethical obligations. In publication of the results of research, the Investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic, or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the subjects who are research subjects.

The benefits, risks, burdens, and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic, or therapeutic method exists.

At the conclusion of the study, every subject entered into the study should be assured of access to the best-proven prophylactic, diagnostic, and therapeutic methods identified by the study.

The physician should fully inform the subject which aspects of the care are related to the research. The refusal of a subject to participate in a study must never interfere with the subject-physician relationship.

In the treatment of a subject, where proven prophylactic, diagnostic, and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the subject, must be free to use unproven or new prophylactic, diagnostic, and therapeutic measures, if in the physician's judgment it offers hope of saving life, reestablishing health, or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases,


new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.


# 16.3 Appendix 3: Commonly Used Corticosteroid Equivalents

| Medication | Prednisone Dose Equivalence |
|--------------------|-----------------------------|
| Prednisone | 1 mg |
| Cortisone | 5 mg |
| Hydrocortisone | 4 mg |
| Prednisolone | 1 mg |
| Methylprednisolone | 0.8 mg |
| Triamcinolone | 0.8 mg |
| Budesonide | 0.25 mg |
| Dexamethasone | 0.16 mg |
| Bethamethasone | 0.16 mg |


# 16.4 Appendix 4: Medication Washout Periods

# WASHOUT TIMES OF MEDICATIONS BASED ON 5 HALF-LIVES

| Medication | Discontinuing Prior to Signing Consent |
|---|---|
| Abatacept (CTLA4Ig) | 24 weeks |
| Alefacept | 12 weeks |
| AMG 623 (blisibimod) | 24 weeks |
| Anifrolumab | 12 weeks |
| Atacicept (TACI-Ig) | 12 weeks |
| Belimumab | 24 weeks |
| Cyclophosphamide | 24 weeks |
| Cyclosporine (except for CSA eye drops) | 4 weeks for oral and 8 weeks for topical |
| Danazol | 4 weeks |
| Dapsone | 4 weeks |
| Eculizumab | 12 weeks |
| Efalizumab | 12 weeks |
| Epratuzumab | 24 weeks |
| Intravenous globulin | 4 weeks |
| Leflunomide | 8 weeks (4 weeks for washout with cholestyramine) |
| Lenalidomide with cholestiramine | 8 weeks |
| Lupuzor | 12 weeks |
| Memantine | 4 weeks |
| Natalizumab | 24 weeks |
| Ocrelizumab | 48 weeks (or 24 weeks with recovery of B cell) |
| Pimecrolimus | 4 weeks |
| Plasmapheresis | 24 weeks |
| Retinoids (oral or topical) | 4 weeks |
| Rituximab | 48 weeks (or 24 weeks with recovery of B cell) |
| Sirolimus | 4 weeks |
| Tacrolimus | 4 weeks |
| Thalidomide | 8 weeks |
| Tocilizumab | 12 weeks |


# 16.5 Appendix 5: BILAG-2004 (Study-Specific Modified Criteria)




# 16.6 Appendix 6: Injection Site Reaction Grading Scale

| Adverse event Injection site reaction | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Definition: A disorder characterized by an intense adverse reaction (usually immunologic) developing at the site of an injection | Tenderness with or without associated symptoms (e.g., warmth, erythema, itching) | Pain;<br>Lipodystrophy;<br>Edema;<br>phlebitis | Ulceration or<br>necrosis;<br>Severe tissue<br>damage;<br>Operative<br>intervention<br>indicated | Life-<br>threatening<br>consequenc<br>es;<br>urgent<br>intervention<br>indicated | Death |
| Pain | Mild pain | Moderate pain;<br>limiting<br>instrumental ADL | Severe pain;<br>limiting self-<br>care ADL | - | - |
| Rash maculopapular/Erythe ma/Induration Definition: A disorder characterized by the presence of macules (flat) and papules (elevated). Also known as morbilliform rash, it is one of the most common cutaneous adverse events, frequently affecting the upper trunk, spreading centripetally, and associated with pruritus. | Macules/papule s covering < 10% BSA with or without symptoms (e.g., pruritus, burning, tightness) Erythema covering < 10% BSA with or without symptoms (e.g., pruritus, burning, tightness) | Macules/papules covering 10% - 30% BSA with or without symptoms (e.g., pruritus, burning, tightness); limiting instrumental ADL; Erythema 30% BSA with or without symptoms (e.g., pruritus, burning, tightness); limiting instrumental ADL | Macules/pap ules covering > 30 % BSA with or without associated symptoms; limiting self-care ADL Erythema covering > 30 % BSA with or without associated symptoms; limiting self-careADL | - | - |

ADL = active daily living


# 16.7 Appendix 7: Opioid Oral Morphine mg Equivalents of Commonly Used Opioids

| Opioid | 30 mg morphine equivalent |
|----------------------|---------------------------|
| butorphanol | 4.3 mg/day |
| codeine | 200 mg/day |
| dihydrocodeine | 120 mg/day |
| fentanyl transdermal | 12.5 mg/day |
| hydrocodone | 30 mg/day |
| hydromorphone | 7.5 mg/day |
| levorphanol tartrate | 2.7 mg/day |
| meperidine HCI | 300 mg/day |
| oxycodone | 20 mg/day |
| oxymorphone | 10 mg/day |
| pentazocine | 81.1 mg/day |
| tapentadol | 75 mg/day |
| tramadol | 300 mg/day |

Note that this list is not comprehensive. If an opioid is being used which is not in this list, please see the appropriate conversion factor below.


## Opioid Oral Morphine Equivalent Conversion Factors<sup>a,b</sup>

| Type of Opioid (strength in units) | MME Conversion Factor |
|---|---|
| Buprenorphine film/table <sup>c</sup> (mg) | 30 |
| Buprenorphine patchd (mcg/hr) | 12.6 |
| Buprenorphine film (mcg) | 0.03 |
| Butorphanol (mg) | 7 |
| Codeine (mg) | 0.15 |
| Dihydrocodeine (mg) | 0.25 |
| Fentanyl buccal or SL tablets, or lozenge/trochee (mcg) | 0.13 |
| Fentanyl film or oral sprayf (mcg) | 0.18 |
| Fentanyl nasal spray <sup>g</sup> (mcg) | 0.16 |
| Fentanyl patchh (mcg) | 7.2 |
| Hydrocodone (mg) | 1 |
| Hydromorphone (mg) | 4 |
| Levorphanol tartrate (mg) | 11 |
| Meperidine hydrochloride (mg) | 0.1 |
| Methadone <sup>i</sup> (mg) | 3 |
| > 0, ≤ 20 | 4 |
| > 20, ≤ 40 | 8 |
| > 40, ≤ 60 | 10 |
| > 60 | 12 |
| Morphine (mg) | 1 |
| Opium (mg) | 1 |
| Oxycodone (mg) | 1.5 |
| Oxymorphone (mg) | 3 |
| Pentazocine (mg) | 0.37 |
| Tapentadol <sup>j</sup> (mg) | 0.4 |
| Tramadol (mg) | 0.1 |

CDC = Centers for Disease Control; CMS = Centers for Medicare and Medicaid Services; FDA = Food and Drug Administration; MAT = Medication Assisted Treatment; MME = morphine mg equivalent; OMS = Overutilization Monitoring System.

The MME conversion factor is intended only for analytic purposes where prescription data is used to calculate daily MME. It is to be used in the formula: Strength per Unit × (Number of Units/Days Supply) × MME conversion factor = MME/Day. This value does not constitute clinical guidance or recommendations for converting patients from one form of opioid analgesic to another. Please consult the manufacturer's full prescribing information for such guidance. Use of this file for the purposes of any clinical decision-making warrants caution.


- National Center for Injury Prevention and Control. CDC compilation of benzodiazepines, muscle relaxants, stimulants, zolpidem, and opioid analgesics with oral morphine mg equivalent conversion factors, 2016 version. Atlanta, GA: Centers for Disease Control and Prevention; 2016. Available at <a href="https://www.cdc.gov/drugoverdose/media/">https://www.cdc.gov/drugoverdose/media/</a>. For more information, send an email to <a href="mailto:Mbohm@cdc.gov">Mbohm@cdc.gov</a>.
- <sup>c</sup> Buprenorphine formulations with a FDA approved indication for MAT are excluded from Medicare's Overutilization Monitoring System's opioid overutilization reporting.
- The MME conversion factor for buprenorphine patches is based on the assumption that 1 mg of parenteral buprenorphine is equivalent to 75 mg of oral morphine and that one patch delivers the dispensed micrograms per hour over a 24 hour day. Example: 5  $\mu$ g/hr buprenorphine patch × 24 hrs = 120  $\mu$ g/day buprenorphine = 0.12 mg/day = 9 mg/day oral MME. In other words, the conversion factor not accounting for days of use would be 9/5 or 1.8.

However, since the buprenorphine patch remains in place for 7 days, we have multiplied the conversion factor by 7 (1.8 × 7 = 12.6). In this example, MME/day for 4 5  $\mu$ g/hr buprenorphine patches dispensed for use over 28 days would work out as follows: Example: 5  $\mu$ g/hr buprenorphine patch × (4 patches/28 days) × 12.6 = 9 MME/day. Please note that because this allowance has been made based on the typical dosage of 1 buprenorphine patch per 7 days, you should first change all Days Supply in your prescription data to follow this standard, i.e., Days Supply for buprenorphine patches = number of patches x 7.

- The MME conversion factor for fentanyl buccal tablets, sublingual tablets, and lozenges/troche is 0.13. This conversion factor should be multiplied by the number of micrograms in a given tablet or lozenge/troche.
- The MME conversion factor for fentanyl film and oral spray is 0.18. This reflects a 40% greater bioavailability for films compared to lozenges/tablets and 38% greater bioavailability for oral sprays compared to lozenges/tablets.
- The MME conversion factor for fentanyl nasal spray is 0.16, which reflects a 20% greater bioavailability for sprays compared to lozenges/tablets.
- The MME conversion factor for fentanyl patches is based on the assumption that 1 mg of parenteral fentanyl is equivalent to 100 mg of oral morphine and that 1 patch delivers the dispensed micrograms per hour over a 24 hour day. Example: 25 μg/hr fentanyl patch × 24 hrs = 600 ug/day fentanyl = 60 mg/day oral morphine mg equivalent.

In other words, the conversion factor not accounting for days of use would be 60/25 or 2.4. However, since the fentanyl patch remains in place for 3 days, we have multiplied the conversion factor by 3 ( $2.4 \times 3 = 7.2$ ). In this example, MME/day for 10 25  $\mu$ g/hr fentanyl patches dispensed for use over 30 days would work out as follows:

Example:  $25 \mu g/hr$  fentanyl patch × (10 patches/30 days) × 7.2 = 60 MME/day. Please note that because this allowance has been made based on the typical dosage of 1 fentanyl patch per 3 days, you should first change all Days Supply in your prescription data to follow this standard, i.e., Days Supply for fentanyl patches = number of patches × 3.

- The CDC MME conversion factor to calculate morphine mg equivalents is 3. CMS uses this conversion factor when analyzing Medicare population opioid use. CMS uses the graduated methadone MME conversion factors to calculate MME within the OMS for identifying and reporting potential opioid overutilizers. https://www.cdc.gov/drugoverdose/pdf/calculating\_total\_daily\_dose-a.pdf.
- Tapentadol is a mu receptor agonist and norepinephrine reuptake inhibitor. Oral MMEs are based on degree of mu-receptor agonist activity, but it is unknown if this drug is associated with overdose in the same dose-dependent manner as observed with medications that are solely mu receptor agonists.


BOS161721 Boston Pharmaceuticals, Inc


# 16.8 Appendix 8: Schedule of Assessments - Phase 1b Multiple Ascending Dose

Table 4. Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Trea | tment | Period | Follov | v-Up | | | | Safet | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28<br>to -1 | 0 | 7<br>(± 1) | 15<br>(± 3) | 30<br>(± 3) | 44<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| | | | | | GENE | RAL AS | SSESS | MENTS | 3 | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | Х | | | | | | | | | | | | | | | |
| Medical history | Х | | | | | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | | | | | |
| SLICC Criteria for SLE | Х | | | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Randomizationc | | Х | | | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | х | | | х | | Х | Х | Х | Х | Х | | | | | |
| | | | - | - | SAFE | TY AS | SESSN | IENTS | | - | | - | - | | - | |
| Full physical exam | Х | Х | | | | | | | | | | | | | | |


<sup>&</sup>lt;sup>a</sup> Screening assessments will be performed over more than 1 visit.

<sup>&</sup>lt;sup>b</sup> Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 4.6.1 for further details.

<sup>&</sup>lt;sup>c</sup> Randomization should occur after patient eligibility has been confirmed by central eligibility review.

Boston Pharmaceuticals, Inc

Clinical Study Protocol: BOS161721-02

BOS161721


Table 4. Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Trea | tment | Period | Follov | v-Up | | | | Safety Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28<br>to -1 | 0 | 7<br>(± 1) | 15<br>(± 3) | 30<br>(± 3) | 44<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| Chest x-rayd | Х | | | | | | | | | | | | | | | |
| C-SSRS | Х | Х | | | | | | Х | | | Х | | | | | |
| AEs and SAEs | | Х | Х | Χ | Х | Х | Χ | Х | Χ | Х | Х | Х | Х | Х | Х | Х |
| 12-lead ECG <sup>e</sup> | Х | Х | | | Х | | | Х | | | | | | | | Х |
| Injection site reaction assessment | | Xf | Х | | х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Targeted physical examination | | | | Х | х | Х | Х | Х | Х | Х | Х | | | Х | Х | Х |
| Vital signs (BP, HR, and temperature) <sup>g</sup> | х | х | | Х | х | Х | Х | Х | Х | Х | Х | | | Х | Х | Х |
| | | | | | EFFIC | ACY A | SSESS | MENT | S | | | | | | | |
| BILAG-2004 Index | Х | Х | | | Х | | Х | Х | Х | Х | Х | | | Х | Х | Х |


<sup>&</sup>lt;sup>d</sup> If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).

<sup>&</sup>lt;sup>e</sup> ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.

<sup>&</sup>lt;sup>f</sup> Injection site reaction assessments to be performed at 2 hours postdose.

<sup>&</sup>lt;sup>9</sup> Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours (±15 minutes) postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, 187, and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection

BOS161721 Boston Pharmaceuticals, Inc


Table 4. Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Trea | tment | Period | Follov | v-Up | | | | Safe | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28<br>to -1 | 0 | 7<br>(± 1) | 15<br>(± 3) | 30<br>(± 3) | 44<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| SLEDAI-2Kh | Х | Χ | | | Χ | | Х | Х | Х | Х | Χ | | | Χ | Х | Χ |
| PGA of disease activity | Х | Х | | | Х | | Х | Х | Х | Х | Х | | | Х | Х | Х |
| ACR-28 joint count | Х | Х | | | Х | | Х | Х | Х | Х | Х | | | Х | Х | Х |
| CLASI | Х | Х | | | Х | | Х | Х | Х | Х | Х | | | Х | Х | Х |
| CCI | | Х | | | Х | | Χ | Х | Χ | Х | Х | | | Х | Х | Х |
| SLICC/ACR<br>Damage Index | | Х | | | | | | | | | Х | | | | | |
| CCI | | Х | | | Х | | Х | Х | Χ | Х | Х | | | Х | Х | Х |
| | • | | | | LABORA | TORY | ASSES | SSMEN | ITS | • | • | • | • | | • | • |
| CD4+ count | Х | Х | | Χ | Х | Х | | Χ | | | Х | | | | | |
| Clinical laboratory<br>assessments<br>(hematology and<br>clinical chemistry) <sup>i</sup> | X | x | | | x | х | х | х | х | х | х | | | X | Х | Х |
| Coomb's test direct <sup>j</sup> | Х | Х | | | Χ | | Х | Х | Х | Х | Χ | | | Х | Х | Х |
| Total IgG and IgM | Х | Х | | Χ | Х | Х | | Х | | | Х | | | | | |
| Plasma CCI | Х | Х | | | Х | | Х | Х | Χ | Х | Х | | | Х | Х | Х |
| Plasma CCI & | | Х | | х | Х | | х | Х | | | Х | | | | | |

<sup>&</sup>lt;sup>h</sup> SLEDAI-2K should be done before randomization and dosing on Day 0 as SLEDAI-2K < 6 is exclusionary


<sup>&</sup>lt;sup>1</sup> Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be non-fasting

<sup>&</sup>lt;sup>j</sup> When clinically indicated for hemolytic anemia

\_\_\_\_

BOS161721 Boston Pharmaceuticals, Inc


Table 4. Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Trea | tment | Period | Follov | v-Up | | | | Safet | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28<br>to -1 | 0 | 7<br>(± 1) | 15<br>(± 3) | 30<br>(± 3) | 44<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| Whole blood for leukocyte immunophenotype | | Х | | Х | х | | Х | Х | | | Х | | | | | |
| ADA <sup>k</sup> | | Х | | Х | Х | | Χ | Χ | | | Χ | | | | | Х |
| nAb <sup>l</sup> | | | | | | | | Χ | | | Х | | | | | |
| pSTAT3 <sup>m</sup> | | Х | | | Х | Х | Χ | Χ | | | | | | | | |
| CCI | | Х | | Χ | | | | Χ | | | Х | | | | | Х |
| CCI | | Х | | | | | | | | | | | | | | |
| CCI | X | X | | | x | | x | x | x | x | x | | | Xn | Xn | Xn |
| CRP | Х | | | | | | | Χ | | | | | | | | Х |
| Serum pregnancy test (women) | Х | | | | | | | | | | | | | | | |


<sup>&</sup>lt;sup>k</sup> Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients, but only assayed (analyzed) if the patient had a positive ADA on Day 90

<sup>&</sup>lt;sup>1</sup> nAb is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90

<sup>&</sup>lt;sup>m</sup> Predose (trough) samples only

<sup>&</sup>lt;sup>n</sup> Antibodies and autoantibodies (CC) will not be analyzed during safety follow-up visits

BOS161721 Boston Pharmaceuticals, Inc


Table 4. Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Trea | tment | Period | Follov | v-Up | | | | Safety Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28<br>to -1 | 0 | 7<br>(± 1) | 15<br>(± 3) | 30<br>(± 3) | 44<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| FSH<br>(postmenopausal<br>women) | Х | | | | | | | | | | | | | | | |
| Urine pregnancy test (women)° | | X | | | X | | Х | Х | Х | Х | X | | | | | Х |
| TB test<br>(QuantiFERON®-TB<br>Gold In-Tube) <sup>d</sup> | Х | | | | | | | | | | | | | | | |
| Serology (hepatitis B and C, HIV-1/2 combination) | X | | | | | | | | | | | | | | | |
| Stool sample <sup>p</sup> | Х | | | | | | | | | | | | | | | |
| Spot urine for protein/creatinine ratio | Х | x | | | x | | Х | Х | Х | Х | Х | | | Х | Х | Х |
| Urinalysis | Х | Χ | | | Х | | Χ | Χ | Х | Х | Х | | | Χ | Χ | Х |
| | | | | | | PK I | Labs | | | | | | | | | |
| Predose | | Χ | | | X | | Χ | Χ | Χ | Χ | Χ | | | | | |
| Predose PK Window | | 60 m | | | ± 3 d | | ±<br>3 d | ±<br>3 d | ±<br>3 d | ±<br>3 d | ± 3 d | | | | | |
| Postdose | | Χq | Χ | Χ | Χq | | | | | | Χq | Χ | Χ | Χ | Χ | Х |


<sup>&</sup>lt;sup>o</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits

<sup>&</sup>lt;sup>p</sup> Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium

<sup>&</sup>lt;sup>q</sup> Postdose samples will be collected at 4, 8, and 24 hours after study drug administration on Days 0, 30, and 180

Table 4. Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | Treatment Period Follow-Up | | | | | | | | | | Safety Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28<br>to -1 | 0 | 7<br>(± 1) | 15<br>(± 3) | 30<br>(± 3) | 44<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| Postdose PK | | 4 h ± | ± 1d | ± 3 d | 4 h ± | | | | | | 4 h ± | ± 3 d | ± 3 d | ± 3 d | ± 3 d | ± 3 d |
| Window | | 30 m | | | 30 m | | | | | | 30 m | | | | | |
| | | 8 h ± | | | 8 h ± | | | | | | 8 h ± | | | | | |
| | | 45 m | | | 45 m | | | | | | 45 m | | | | | |
| | | 24 h ± | | | 24 h ± | | | | | | 24h ± | | | | | |
| | | 60 m | | | 60 m | | | | | | 60 m | | | | | |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; APL = antiphospholipid;
BILAG = British Isles Lupus Assessment Group; BP = blood pressure; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CLASI = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CLASI = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CLASI = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CLASI = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CLASI = FOR = FOR = C-PSSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CLASI = FOR = ECG = electrocardiogram; CLASI = CLASI = CLASI = CLASI = CLASI = CLASI = Adverse event; CLASI = CLASI = Adverse event; CLASI = Adverse event; CLASI = Adverse event; CLASI = CLASI = Adverse event; CLASI = CLASI = Adverse event; CLASI = Adverse ev


#### 16.9 Appendix 9: Protocol Summary of Changes

The COVID-19 pandemic, caused by the SARS-CoV-2 virus, has necessitated social distancing and shelter-in-place type practices and limited transportation globally. A contingency plan was implemented in anticipation of disruptions to study visits and study assessments. This amendment summarizes the measures implemented during the COVID-19 pandemic to protect patient safety and data integrity.

- Safety oversight: In case a patient cannot return to the study site for the scheduled visit, the site staff will contact the patient remotely for safety follow up, for example, via telephone or video conferencing.
- Central Laboratory: In the case that there are courier issues that will prevent the
  protocol-required laboratory specimens to be sent to the study core laboratory, the
  site should have the safety laboratory specimens (Table 2: Hematology, Chemistry,
  and Urinalysis) sent to their local laboratory for analysis and review by the study
  physician.
- Investigational Product Dosing: In cases when dosing cannot be performed during the protocol-designated windows, the Investigator should discuss each case with the Sponsor to determine whether it is a missed visit or whether the dosing can be performed outside protocol windows (as a protocol deviation). A minimum of 2 weeks must be maintained between consecutive doses. Patients who miss more than 2 doses of the study drug (whether consecutive or not) will be discontinued from the study and will undergo assessments as outlined in Section 5.5 (Premature Discontinuation).

Additional changes in this amendment include:

- 1. Sample size recalculation based on data from the Ustekinumab Phase 2 study in SLE.
- 2. Revisions to secondary and exploratory endpoints based on precedence in other successful clinical trials and to account for SLE disease heterogeneity.
- 3. Additional options for acceptable contraception methods.

Significant changes are described in the table below. Changed text is displayed for the first major occurrence only. Deleted text is presented in strikethrough format, and added text is presented in bold format.

| Section | Description of Changes | Rationale |
|---------|------------------------------------------------|----------------|
| Global | Replace: | Administrative |
| | Protocol Date and Version: 23 July 2019; V6.0 | |
| | With: | |
| | Protocol Date and Version: 30 April 2020; V7.0 | |
| Global | Change: | Administrative |


| Section | Description of Changes | Rationale |
|---|---|---|
| | Changed Version number from V6.0 (Amendment 5) to V7.0 (Amendment 6) and Version date from 23 July 2019 to 30 April 2020. | |
| Global | Made administrative and editorial (formatting, typographical, and grammatical) updates. | Administrative |
| CLINICAL<br>PROTOCOL<br>APPROVAL FORM | Replace: Name and Title PPD , MD, PhD Chief Medical Officer Boston Pharmaceuticals With: Name and Title PPD , MD, PhD Chief Medical Officer Boston Pharmaceuticals | New CMO. |
| CLINICAL<br>PROTOCOL<br>APPROVAL FORM | Replace: Name and Title PPD , PhD Senior Vice President Clinical Development and Head of Clinical Operations Boston Pharmaceuticals With: Name and Title PPD , MD Vice President Clinical Development Boston Pharmaceuticals | New clinical lead for the program. |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>Phase 2,<br>Secondary | Replace: Results and changes from baseline in: With: Changes and percent changes from baseline in: | SLE is a very heterogeneous disease. As a result, baseline data could vary considerably from patient to patient. Percent change from baseline enables |


| Section | Description of Changes | Rationale |
|---|---|---|
| Endpoints, Bullet 2 (sub-bullet 2) | | comparison between treatment arms despite baseline variability. |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>Phase 2,<br>Secondary<br>Endpoints, Bullet 2<br>(sub-bullet 2) | Replace: The Results and changes from baseline in: CLASI With: The Changes and percent changes from baseline in: CLASI PGA | PGA is added as an important disease activity score in SLE. |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>Phase 2,<br>Secondary<br>Endpoints, Bullet 6 | Remove: Time to first SRI-4 response | This endpoint is removed since the SRI-4 response is not always stable and could disappear from one visit to next. |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>Phase 2,<br>Exploratory<br>Endpoints | Insert: CCI CCI CCI CCI CCI CCI CCI C | |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>phase 2,<br>Exploratory<br>Endpoints, second<br>row, second<br>column, Bullet 2 | Replace: | CCI |
| INTRODUCTION<br>AND RATIONALE,<br>Section 1.2.5,<br>Potential Risks,<br>Sub-section | Replace: Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells, patients with a CD4+ count < 500 cell/mm³ were | The text is made consistent with the revised eligibility criteria for CD4+ count in POC. |


| Section | Description of Changes | Rationale |
|---|---|---|
| 1.2.5.4, Infections, Paragraph 7. | excluded from the Phase 1 SAD study (BOS161721-01), and CD4+ < 350 cells/mm³ will be excluded from the MAD/POC parts of the study. With: Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells, patients with a CD4+ count < 500 cell/mm³ were excluded from the phase 1 SAD study (BOS161721-01). Patients with CD4+ count < 350 cells/mm³ and CD4+ count < 150 cells/mm³ will be excluded from the MAD and POC parts of the study, respectively. | |
| STUDY OBJECTIVES AND ENDPOINTS, Section 2.2, phase 2 Proof of Concept, Secondary Endpoints, Bullet 2. | Replace: Results and changes from baseline in: With: Changes and percent changes from baseline in: | SLE is a very heterogeneous disease. As a result, baseline data could vary considerably from patient to patient. Percent change from baseline enables comparison between treatment arms despite baseline variability. |
| STUDY OBJECTIVES AND ENDPOINTS, Section 2.2, phase 2 Proof of Concept, Secondary Endpoints, Bullet 2. | Replace: The Results and changes from baseline in: CLASI With: The Changes and percent changes from baseline in: CLASI PGA | PGA is added as an important disease activity score in SLE. |
| STUDY OBJECTIVES AND ENDPOINTS, Section 2.2, phase 2 Proof of Concept, Secondary Endpoints, Bullet 6. | Remove: Time to first SRI-4 response | This endpoint is removed since the SRI-4 response is not always stable and could disappear from one visit to next. |


#### BOS161721


| Section | Description of Changes | Rationale |
|---|---|---|
| STUDY OBJECTIVES AND ENDPOINTS, Section 2.2, phase 2 Proof of Concept, Exploratory Endpoints | Insert: CCI CCI CCI CCI CCI CCI CCI C | CCI |
| STUDY OBJECTIVES AND ENDPOINTS, Section 2.2, phase 2 Proof of Concept, Exploratory Endpoints, second row, second column, Bullet 2 | Replace: CCI | CCI |
| STUDY PLAN,<br>Section 3.1.1,<br>Multiple Ascending<br>Dose Phase 1b, | Replace: All doses selected for the MAD part of the study are projected not to exceed the mean exposure of that achieved in the SAD study. With: All doses selected for the MAD part of the study are projected not to exceed the mean exposure of that achieved at the highest dose in the SAD study. | Clarification is made as to the approach to dose selection. |
| STUDY PLAN,<br>Section 3.1.2.2,<br>POC Study Design | Replace: For the POC part of the study, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio. With: For the POC part of the study, approximately 110 additional patients will be randomized to active or placebo groups in a 2:1 ratio. | Efficacy data from a Phase 2 SLE study of SRI-4 response to Ustekinumab, which has a partially overlapping mechanism of action on T cells, became available <sup>51</sup> and was therefore used to reassess power calculations in this study of BOS-161721 of SRI-4 response in SLE. Ustekinumab produced a |


| Section | Description of Changes | Rationale |
|---|---|---|
| | | statistically significant difference in SRI-4 response in favor of Ustekinumab (62% Ustekinumab vs. 33% placebo) with 102 patients. Therefore, sample size was reduced in BOS161721-02 from 156 to 96 evaluable patients. |
| STUDY PLAN, | Replace: | Efficacy data from a |
| Section 3.2, Randonization and | Phase 2 156* 2:1 | Phase 2 SLE study of SRI-4 response to |
| Blinding | With: | Ustekinumab, which has a partially overlapping |
| CTHDY DI ANI | Phase 2 Approximately 110 2:1 | mechanism of action on T cells, became available <sup>51</sup> and was therefore used to reassess power calculations in this study of BOS-161721 of SRI-4 response in SLE. Ustekinumab produced a statistically significant difference in SRI-4 response in favor of Ustekinumab (62% Ustekinumab vs. 33% placebo) with 102 patients. Therefore, sample size was reduced in BOS161721-02 from 156 to 96 evaluable patients. |
| STUDY PLAN,<br>Section 3.4,<br>Schedule of<br>Assessments | Replace: Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 187 and 195). With: Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours (± 15 minutes) postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 187 and 195). | Flexible language is introduced for the timing of the vital signs. |
| STUDY PLAN,<br>Section 4.2,<br>Number of Patients | Replace: Approximately 186 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, | Sample size<br>re-calculation was<br>performed based on<br>recent data from the |


| Section | Description of Changes | Rationale |
|---|---|---|
| | which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD Phase 1b portion, and approximately 156 additional patients will be randomized in the POC Phase 2 portion. Note that approximately 24 dropouts are assumed. With: | Ustekinumab phase 2<br>study. Please see<br>Section 8.1. |
| | Approximately 140 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD phase 1b portion, and approximately 110 additional patients will be randomized in the POC phase 2 portion. Note that approximately 14 dropouts are assumed in the POC phase 2 portion. | |
| STUDY PLAN, | Replace: | As many patients with |
| Section 4.7.2,<br>Contraception | Patients must agree to either complete abstinence, defined as a complete avoidance of heterosexual activity, or the use of 2 methods of highly effective contraception from the following: • Male condoms with spermicide • Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug • IUDs, such as ParaGard® • Vasectomy • Note: Women who are abstinent while participating in the study must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the patient chooses to forego complete abstinence • Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. | SLE are unable to tolerate hormonal contraception, additional effective methods of contraception (diaphragm with spermicide, cervical cap with spermicide and hormonal patches) were introduced to provide more flexibility for study participants. |
| | However, WOCBP must still undergo pregnancy testing With: | |


| Section | Description of Changes | Rationale |
|---|---|---|
| | Patients must agree to either complete abstinence, defined as a complete avoidance of heterosexual activity, or the use of 2 methods of effective contraception from the following: | |
| | Male condoms with spermicide | |
| | Diaphragm with spermicide | |
| | Cervical cap with spermicide | |
| | Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, patches, and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug | |
| | <ul> <li>IUDs, such as ParaGard®</li> </ul> | |
| | <ul> <li>Vasectomy</li> </ul> | |
| | Note: Women who are abstinent while participating in the study must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the patient chooses to forego complete abstinence | |
| | <ul> <li>Azoospermic men and WOCBP who are<br/>continuously not heterosexually active are<br/>exempt from contraceptive requirements.<br/>However, WOCBP must still undergo<br/>pregnancy testing</li> </ul> | |
| STUDY PLAN,<br>Section 5.2,<br>Enrollment/Random<br>ization and Day 0<br>Treatment | <ul> <li>Replace:</li> <li>Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours postdose on Day 0)</li> <li>With:</li> <li>Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours [± 15 minutes] postdose on Day 0)</li> </ul> | Flexible language is introduced for the timing of the vital signs. |
| STUDY PLAN, Section 5.6, Contingency Plans During the COVID-19 Pandemic | <ul> <li>Safety oversight: In case a patient cannot return to the study site for the scheduled visit, the site staff will contact the patient remotely for safety follow up, for example, via telephone or video conferencing.</li> <li>Central Laboratory: In the case there are courier issues that will prevent the protocol-required</li> </ul> | During the COVID-19 pandemic, due to social distancing and shelter-in-place type practices and limitations in transportation, measures were implemented to protect patient safety and data |
| | laboratory specimens to be sent to the study core laboratory, the site should have the safety | integrity. |


| Section | Description of Changes | Rationale |
|---|---|---|
| | laboratory speciments (Table 2: Hematology, Chemistry, and Urinalysis) sent to their local laboratory for analysis and review by the study physician. | |
| | Investigational Product Dosing: In cases when dosing cannot be performed during the protocol-designated windows, the Investigator should discuss each case with the Sponsor to determine whether it is a missed visit or whether the dosing can be performed outside protocol windows (as a protocol deviation). A minimum of 2 weeks must be maintained between consecutive doses. Patients who miss more than 2 doses of the study drug (whether consecutive or not) will be discontinued from the study and will undergo assessments as outlined in Section 5.5 (Premature Discontinuation). | |
| ASSESSMENTS,<br>Section 6.2.3,<br>Vital Signs | Replace: Vital signs will be assessed on Day 0 at predose and at Day 0, 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). | Flexible language is introduced for the timing of the vital signs. |
| | With: Vital signs will be assessed on Day 0 at predose and at Day 0, 1 and 2 hours (± 15 minutes) postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). | |
| ASSESSMENTS,<br>Section 6.3.5,<br>CLASI Response,<br>Paragraph 1. | Replace: This assessment will be applied to all patients as all are required to have cutaneous disease activity. With: This assessment will be applied to all patients who have cutaneous disease activity. | Inclusion criteria could be met without presence of mucocutaneous disease. |
| STATISTICS,<br>Section 8.1,<br>Sample Size | Replace: The sample size in the Phase 2 portion is based on the primary endpoint, SRI-4 Response at Day 210. Approximately 156 additional patients will be randomized in a 2:1 ratio to BOS161721 versus placebo to achieve 132 evaluable patients in the FAS. This assumes 24 patients will drop prior to having received treatment and an evaluable post-baseline efficacy measure. Enrollment and randomization will be monitored in a blinded fashion and increased if needed to ensure at least 132 patients are randomized into the FAS. A total of 132 patients randomized provides more than 80% power to detect a treatment difference of 25% in SRI-4 response rates at Day 210, based on a targeted 2-sided significance level of 10% and | Efficacy data from a Phase 2 SLE study of SRI-4 response to Ustekinumab, which has a partially overlapping mechanism of action on T cells, became available <sup>51</sup> and was therefore used to reassess power calculations in this study of BOS-161721 of SRI-4 response in SLE. Ustekinumab produced a statistically significant difference in SRI-4 response in favor of |


| Section | Description of Changes | Rationale |
|---|---|---|
| | using a 2-sided Pearson's chi-squared test. This assumes of a response rate of 65% for BOS161721 and 40% for placebo, where missing data at Day 210 is carried forward from most recent non-missing result and patients are treated as a non-responder if a prohibited medication defined as a medication failure occurs. With: | Ustekinumab (62%<br>Ustekinumab vs. 33%<br>placebo) with 102<br>patients. Therefore,<br>sample size was reduced<br>in BOS161721-02 from<br>156 to 96 evaluable<br>patients. |
| | The sample size in the phase 2 portion is based on the primary endpoint, SRI-4 Response at Day 210. Based on efficacy data from a recently completed study with Ustekinumab, where the primary endpoint was also SRI-4, the sample size in the phase 2 part of the BOS161721-02 study is set at 96 evaluable patients. In the Ustekinumab study of 102 patients, a statistically significant difference in SRI-4 response was shown in favor of Ustekinumab (62% of Ustekinumab treated patients achieved SRI-4 response vs. 33% in patients receiving placebo). The Ustekinumab phase 2 study is an appropriate comparator to BOS161721-02 because both studies share the same primary endpoint of SRI-4 response and BOS161721 and Ustekinumab have overlapping mechanisms of action (T follicular helper and Th17 cell biology). | |
| | Approximately 110 additional patients will be randomized in a 2:1 ratio to BOS161721 versus placebo to achieve approximately 96 evaluable patients in the FAS of the phase 2 portion. This assumes 14 patients will drop prior to having received treatment or having completed a post-baseline efficacy measure. Enrollment and randomization will be monitored in a blinded fashion and may be increased if needed to ensure at least 96 evaluable patients are randomized into the FAS. | |
| | A total of 96 evaluable patients randomized provides 80% power to detect a treatment difference of 29% in SRI-4 response rates at Day 210, based on a targeted 2-sided significance level of 10% and using a 2-sided Pearson's chi-squared test. This assumes a response rate of 62% for BOS161721 and 33% for placebo. | |
| STATISTICS,<br>Section 8.2.1,<br>Analysis<br>Populations,<br>Paragraph 1 and 3 | Inserted:<br>(partial or complete) | Words partial or complete are added for further clarity. |
| STATISTICS,<br>Section 8.2.3,<br>Primary Efficacy | Replace: The proportion of patients who achieve a SRI-4 response at Day 210 will be assessed via Pearson's chi-squared analysis. The primary efficacy endpoint | Flexible language is introduced to perform additional analyses or apply additional |


| Section | Description of Changes | Rationale |
|---|---|---|
| Endpoint(s),<br>Paragraph 1 and 2. | will be analyzed using the FAS and if needed repeated in the PP analysis set. Missing values will be addressed by employing a last observation carried forward (LOCF) analysis. Other imputation methods may be employed as a sensitivity analysis and will be described in the SAP. Additional analyses exploring impact of baseline factors such as baseline disease severity, race, and other characteristics may be performed. With: | impuation methodology based on emerging data. |
| | The proportion of patients who achieve a SRI-4 response at Day 210 will be assessed via Pearson's chi-squared analysis. The primary efficacy endpoint will be analyzed using the FAS and if needed repeated in the PP analysis set. Missing values will be addressed by employing a last observation carried forward (LOCF) analysis. Other imputation methods may be employed as a sensitivity analysis and will be described in the SAP. Analyses based on observed values may also be performed. Exploratory subgroup analyses assessing impact of baseline factors such as baseline disease severity, background therapy, race, geography, baseline serologic activity, and other characteristics may be | |
| | performed. Additional exploratory analyses of disease activity endpoints may be performed based on emerging data. | |
| APPENDICIES,<br>Section 16.8,<br>Appendix 8,<br>Table 4 Schedule<br>of Assessments -<br>Phase 1b Multiple<br>Assceding Dose | Replace: Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, 187, and 195). With: | Flexible language is introduced for the timing of the vital signs. |
| | Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours (±15 minutes) postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, 187, and 195). | |




#### **Certificate Of Completion**

Envelope Id: PPD

Subject: Please DocuSign: BOS161721-02\_Protocol\_Amendment 6\_V 7 0\_Clean\_30Apr2020.docx

Source Envelope:

Document Pages: 130 Certificate Pages: 5

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

**Envelope Originator:** 

PPD

PPD

PPD

PPD PPD

#### **Record Tracking**

Status: Original

5/5/2020 1:46:10 PM

Holder: PPD

Signatures: 3

Initials: 0

Location: DocuSign

#### **Signer Events**

PPD

Security Level: Email, Account Authentication

(Required)

**Signature** 

PPD

Signature Adoption: Pre-selected Style

Signature ID:

Using IP Address: PPD Signed using mobile

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 5/6/2020 7:06:37 AM

ID: PPD

PPD

Security Level: Email, Account Authentication

(Required)

PPD

Signature Adoption: Pre-selected Style

Signature ID:

PPD

Using IP Address: PPD

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 5/6/2020 9:57:01 AM

ID: PPD

**Timestamp** 

Sent: 5/5/2020 1:50:48 PM Viewed: 5/6/2020 7:06:37 AM Signed: 5/6/2020 7:07:11 AM

Sent: 5/5/2020 1:50:48 PM Viewed: 5/6/2020 9:57:01 AM Signed: 5/6/2020 9:57:24 AM

**Signer Events Signature Timestamp** PPD Sent: 5/5/2020 1:50:48 PM PPD Viewed: 5/5/2020 3:46:16 PM Security Level: Email, Account Authentication (Required) Signed: 5/5/2020 3:46:47 PM Signature Adoption: Pre-selected Style Signature ID: PPD Using IP Address: PPD

> With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

# Electronic Record and Signature Disclosure: Accepted: 5/5/2020 3:46:16 PM ID: PPD

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Summary Events Envelope Sent Certified Delivered Signing Complete Completed | Status Hashed/Encrypted Security Checked Security Checked Security Checked | Timestamps 5/5/2020 1:50:48 PM 5/6/2020 9:57:01 AM 5/6/2020 9:57:24 AM 5/6/2020 9:57:24 AM |
| Envelope Sent Certified Delivered Signing Complete | Hashed/Encrypted Security Checked Security Checked | 5/5/2020 1:50:48 PM<br>5/6/2020 9:57:01 AM<br>5/6/2020 9:57:24 AM |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, MMS Holdings Inc. (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact MMS Holdings Inc.:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

#### To advise MMS Holdings Inc. of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at PPD and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

#### To request paper copies from MMS Holdings Inc.

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to PPD and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with MMS Holdings Inc.

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to PPD and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| required hard ware and software | |
|---|---|
| Operating Systems: | Windows2000? or WindowsXP? |
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy<br>Server must enable HTTP 1.1 settings via<br>proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify MMS Holdings Inc. as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by MMS Holdings Inc. during the course of my relationship with you.

BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 23 July 2019; V6.0



# A RANDOMIZED DOUBLE-BLIND PHASE 1b/2 COMBINED STAGGERED MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF LIMITED STANDARD OF CARE

**SPONSOR** Boston Pharmaceuticals, Inc.

55 Cambridge Parkway, Suite 400

Cambridge, MA 02142

United States of America (USA)

INVESTIGATIONAL COMPOUND: BOS161721

PROTOCOL NUMBER: BOS161721-02

PHASE Phase 1b/2

INVESTIGATIONAL NEW DRUG (IND) 131796

**NUMBER:** 


**VERSION NUMBER:** V6.0 (Amendment 5)

VERSION DATE: 23 July 2019


## CLINICAL PROTOCOL APPROVAL FORM

| Protocol Title: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care | |
|---|---|
| Study Number: | BOS161721-02 |
| Version | Date |
| Original Protocol | 06 October 2017 |
| Protocol Version 2.0 (Amendment 1) | 14 November 2017 |
| Protocol Version 3.0 (Amendment 2) | 21 March 2018 |
| Protocol Version 4.0 (Amendment 3) 27 July 2018 | |
| Protocol Version 5.0 (Amendment 4) 23 January 2019 | |
| Protocol Version 6.0 (Amendment 5) | 23 July 2019 |

This study protocol was subject to critical review and has been approved by sponsor. The information contained in this protocol is consistent with:

- The current risk-benefit evaluation of the investigational product.
- The moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (APPENDIX 2), and principles of Good Clinical Practices (GCP) as described in 21 Code of Federal Regulations (CFR) parts 50, 54, 56 and 312 and according to applicable local requirements.

The investigator will be supplied with details of any significant or new findings, including adverse events, relating to treatment with the investigational product.

I agree with these statements and indicate my approval by signature for this protocol:

| Name and Title | Signature and Date |
|---|---|
| PPD , MD, PhD Chief Medical Officer | PPD |
| Boston Pharmaceuticals | |
| PPD , PhD Senior Vice President Clinical Development and Head of Clinical Operations Boston Pharmaceuticals | PPD ( |
| PPD Clinical Operations Lead Boston Pharmaceuticals | PPD |


#### BOS161721-02

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

#### CONFIDENTIALITY AND INVESTIGATOR STATEMENT

The information contained in this protocol and all other information relevant to BOS161721 are the confidential and proprietary information of Boston Pharmaceuticals, Inc., and except as may be required by federal, state, or local laws or regulation, may not be disclosed to others without prior written permission of Boston Pharmaceuticals, Inc.

I have read the protocol (Version 6.0, dated 23 July 2019), including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described. I will conduct this study as outlined herein, in accordance with the regulations stated in the Federal Code of Regulations for Good Clinical Practices and International Council for Harmonisation (ICH) guidelines, and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and any amendments, and access to all information provided by Boston Pharmaceuticals, Inc., or specified designees. I will discuss the material with them to ensure that they are fully informed about BOS161721 and the study.

| Principal Investigator Name (printed) | | Signature |
|---------------------------------------|-------------|-----------|
| Date | Site Number | |


# PROTOCOL SUMMARY

| Title: | A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care |
|---|---|
| Indication | Adults with moderately to severely active SLE |
| Background and Rationale | SLE is a chronic systemic autoimmune disease with considerable heterogeneity in clinical manifestations and disease course. There is evidence that B- and T-cells are critical to the development of the disease, and that T-cell-derived cytokines such as interleukin-21 (IL-21) are involved in the SLE-associated inflammatory pathological response. |
| | BOS161721 is a humanized immunoglobulin G1 (IgG1) triple mutation monoclonal antibody (mAb) intended to have an extended terminal elimination half-life (t½) that selectively binds to and neutralizes IL-21, which acts on multiple cell types that drive inflammation and autoimmunity. <i>In vivo</i> , BOS161721 inhibits T-cell dependent antigen responses of B-cells and is being developed as a potential treatment for adults with moderately to severely active SLE. |
| | Nonclinical studies have evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), pharmacokinetics (PK), and immunogenicity of BOS161721 administered intravenously (IV) and subcutaneously (SC). The no observed adverse effect level (NOAEL) in Cynomolgus monkeys was determined to be 100 mg/kg (SC and IV), the highest dose tested. There were no injection site reactions in animals dosed subcutaneously. |
| | In a Phase 1 single ascending dose (SAD) study, BOS161721 was administered IV and SC to healthy male and female adult subjects. This double-blind, placebo-controlled study evaluated 8 ascending dose levels (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) for safety, tolerability, PK, PD and immunogenicity. Overall, there were no clinically significant safety or tolerability findings from this study. |
| | Results from the Phase 1 SAD study informed the dose regimens used for the multiple ascending doses (MAD) Phase 1b portion of this trial. The MAD portion will involve 3 cohorts. The Phase 2 portion will be a proof of concept (POC) part, where dose selection will be based on the data monitoring committee (DMC) and sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD portion of 30 patients treated with BOS161721/placebo. The purpose of the study is to establish a safe and effective dosage for adult patients with moderately to severely active SLE. |


BOS161721 Boston Pharmaceuticals, Inc.


# **Objectives and Endpoints:**

### **MAD Phase 1b**

#### **OBJECTIVES ENDPOINTS** Primary To assess safety, tolerability, and Safety Endpoints immunogenicity of repeat doses of Incidence and severity of adverse events BOS161721 (20, 60, and 120 mg) (AEs) and serious adverse events (SAEs), administered SC in adult patients related AEs, AEs leading to study drug with moderately to severely active discontinuation, AEs by severity and SLE on limited background relatedness standard of care treatment, in order Injection site reactions to estimate the optimal dose. Columbia Suicide Severity Rating Scale 12-lead electrocardiograms (ECGs) parameter results at each visit and change from baseline Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline Clinical laboratory results and change from baseline Physical examinations changes from baseline Anti-drug antibodies (ADAs) Study drug exposure/compliance **Secondary** To characterize the PK of Pharmacokinetic Endpoints BOS161721 and select the optimal BOS161721 concentration by visit and time dose of BOS161721 based on point safety, PK, and PD effects in Maximum observed concentration (C<sub>max</sub>), patients with moderately to first time to maximum concentration (T<sub>max</sub>), severely active SLE. area under the concentration-time curve (AUC), t<sub>1/2</sub>, systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>) Pharmacodynamic Endpoints Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit





# **POC Phase 2**

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To demonstrate a superior effect of<br>BOS161721 at the chosen dose<br>compared with placebo for<br>response on the SLE Responder<br>Index 4 (SRI-4) | <ul> <li>Primary Efficacy Endpoint</li> <li>The proportion of patients with a SRI-4 response at Day 210 (see Section 6.3.4.1)</li> </ul> |
| Secondary | |
| To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment Sofetice Sofetice To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment | <ul> <li>The proportion of patients with: <ul> <li>SRI-4 response at each visit</li> <li>SRI-5 and SRI-6 response at each visit (Section 6.3.4.2)</li> <li>a sustained reduction from baseline of oral corticosteroid (CS) (≤ 7.5 mg/day and &lt; Day 0 dose) between Day 150 and Day 210</li> <li>new or recurrent BILAG flares (≥ 1 qualifying BILAG A or &gt; 1 qualifying BILAG B) through Day 210</li> <li>PGA worsening</li> <li>a BICLA response</li> <li>a CLASI response</li> <li>medication failures</li> </ul> </li> <li>Results and changes from baseline in: <ul> <li>CLASI</li> <li>Total number of swollen joints, tender joints, and active joints (swelling and tenderness in the same joint) in the ACR-28 joint count</li> <li>SLEDAI-2K</li> <li>SLICC/ACR damage index</li> </ul> </li> <li>Time to medication failure</li> <li>Group mean percent reduction in corticosteroid administration from baseline Day 0 dose through Day 210 in patients receiving ≥ 7.5 mg/day prednisone equivalent at Day 0</li> <li>Duration of longest SRI-4 response</li> <li>Time to first SRI-4 response</li> <li>Time to first SRI-4 response</li> <li>Time to first BILAG flare (≥ 1 new or recurrent BILAG B) relative to baseline through Day 210</li> </ul> |
| Safety | |
| To assess safety and tolerability of<br>repeat doses of BOS161721 at the<br>chosen dose administered SC in | Safety Endpoints Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), |


BOS161721 Boston Pharmaceuticals, Inc.




#### **Study Design:**

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of multiple SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, eligible patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly. The trial will consist of 2 double-blinded portions: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

The MAD Phase 1b portion of the study design will consist of 3 cohorts, with


Cohort 1 containing 6 patients, where 5 of these patients will receive BOS161721 (active), and 1 will receive placebo. Cohorts 2 and 3 will each contain 12 patients, including 9 active and 3 placebo patients. Dose selection for each cohort is based on 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. Each of the 3 doses (20, 60, and 120 mg) selected for the MAD portion are projected not to exceed the mean exposure of that achieved in the SAD study following the single 240 mg SC dose. Each patient may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

The MAD portion design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after the DMC evaluates the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after the DMC evaluation of the safety and tolerability data from Cohort 2 and Cohort 1. Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. This dose will not exceed doses tested during the MAD portion.

For the POC portion, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio. As in the MAD portion, each patient in the POC portion may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

A maximum stable (for at least 6 weeks prior to Day 0) daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study. One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 120. Tapering of steroids during the course of the study will be highly encouraged and should be evaluated during the protocol-allowed tapering windows (Day 0 through Day 150) with the target of achieving a CS daily dose of  $\leq 7.5$  mg and < Day 0 dose between Day 150 and Day 210. Between Day 150 and Day 210, oral CS doses must be held constant due to the Day 210 endpoint evaluations.

DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.


# Main Criteria for Inclusion and Exclusion

#### **Inclusion Criteria:**

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion OR Lupus nephritis as the sole clinical criterion in the presence of antinuclear antibodies [ANA] or anti- double-stranded deoxyribonucleic acid [dsDNA] antibodies), either sequentially or simultaneously
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
- 5. At screening, the total SLEDAI-2K score must be  $\geq 8$ , including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

- 6. A clinical SLEDAI-2K score of  $\geq 6$  at screening at Day 0. Clinical SLEDAI-2K score is defined as follows:
  - a. Contains points from arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, or vasculitis
  - b. Excludes parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.


7. Patients must have at least 1 qualifying A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:

- a. BILAG A or B score in the mucocutaneous body system. If a BILAG B score is due to BILAG number 6, mild skin eruption, the CLASI activity score including erythema and scale/hypertrophy must be ≥ 3 excluding points from mucosal ulcers and alopecia.
- b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 4.4

Note: Hips, shoulders, back, neck, and temporomandibular joints do not count towards the total number of joints with active synovitis.

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in at least 1 other body system for a total of 2 "B" BILAG body system scores.

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to Day 0) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. If AZA, myocophenolate mofetil, mycophenolic acid, hydroxychloroquine, or MTX were discontinued prior to screening, the washout period must be ≥ 12 weeks.
  - c. Corticosteroids (prednisone or prednisone-equivalent) at a stable dose of up to 30 mg/day for at least 6 weeks prior to Day 0 (see APPENDIX 3)
    - i. For patients whose only SLE treatment is CSs, the stable CS dose must be  $\geq 10$  mg/day for at least 6 weeks prior to Day 0 and no more than 30 mg/day at the time of randomization.
    - ii. Topical steroids may be used, but the dose must be stable for at least 6 weeks prior to Day 0. PRN topical steroids are not permitted.
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and


### contraception):

- a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
- b. Must not be breastfeeding
- c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

#### **Exclusion Criteria**

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic sclerosis, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed
- 5. Active or unstable lupus neuropsychiatric manifestations, including but


not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed

- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator or the sponsor or their designee, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count  $< 150/\mu$ L at screening
- 16. Platelets < 50,000/mm<sup>3</sup> (50  $\times$  10<sup>9</sup>/L) or < 35,000/ mm<sup>3</sup> (35  $\times$  10<sup>9</sup>/L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation
- 20. Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) > 2 × the upper limit of normal (ULN) at screening, unless explicitly related to lupus based on the investigator's judgment


- 21. Creatinine kinase (CK) > 3.0 × ULN at screening unless related to lupus myositis
- 22. Total bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator or the sponsor or sponsor's designee, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic mAb (eg, IgG protein) or molecules made of components of mAbs
- 25. History substance and/or alcohol abuse, or dependence within the past 1 year, at the investigator's judgment
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision)
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, sponsor or sponsor's designee, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 on the C-SSRS
- 31. Current or pending incarceration
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness
- 33. Currently taking a total daily dose of > 30 mg morphine or morphine equivalent (see APPENDIX 7)
- 34. Body mass index (BMI)  $\geq$  40.0

# Statistical Considerations

Below is a summary of the statistical methods. Further details can be found in Section 8.

Two analyses are planned: 1) an interim analysis to select the POC dose based on the MAD data, and 2) a final analysis at study completion.


Additionally, DMC safety analyses will be performed for each MAD cohort and throughout the POC to monitor patient safety as described in the DMC charter. An additional analysis may be performed for the MAD portion of the study when all MAD patients have completed the safety follow-up, or withdrawn from the study, and prior to the final analysis. Data from the POC part of the study will be excluded from this additional analysis.

Unless stated otherwise, statistical testing will only be performed on the POC data and will be done using 2-sided overall alpha of 0.10. Data will be summarized descriptively by treatment and overall for each study phase. For the MAD portion, BOS161721 will be summarized overall and by each dose level and placebo patients from each cohort will be combined.

The descriptive summaries for the categorical data will include number and percentage. The descriptive summaries for the continuous data will include number, mean, median, standard deviations (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, median, and maximum. Counts, medians, 25<sup>th</sup> and 75<sup>th</sup> percentiles, and standard error will be presented for time-to-event data.

All safety analyses will be performed using the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. All efficacy analyses will be performed using the full analysis set (FAS), defined as all patients who receive at least 1 dose of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. Select efficacy analyses may also be performed on the per protocol (PP) set.

Binary efficacy endpoints, including the primary efficacy endpoint, will be assessed via Pearson's chi-squared analysis.

Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) when applicable, adjusting for the baseline value. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test.

Adverse event data will be coded to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be summarized, based on coded terms, using frequency and percentage of patients. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters, will be summarized at each individual visit.


# **TABLE OF CONTENTS**

| CLINICAL PROTOCOL APPROVAL FORM | 2 |
|----------------------------------------------------|--------|
| CONFIDENTIALITY AND INVESTIGATOR STATEMEN | Τ3 |
| PROTOCOL SUMMARY | |
| TABLE OF CONTENTS | 16 |
| LIST OF IN-TEXT TABLES | 19 |
| LIST OF IN-TEXT FIGURES | 20 |
| LIST OF ABBREVIATIONS | 21 |
| 1. INTRODUCTION AND RATIONALE | 25 |
| 1.1 Indication | 25 |
| 1.2 Background and Rationale | 25 |
| 1.2.1 Overview of the Disease State | 25 |
| 1.2.2 BOS161721 Development | 25 |
| 1.2.2.1 Interleukin-21 | 26 |
| 1.2.2.2 Preclinical Studies | 27 |
| 1.2.2.3 Clinical Studies | 28 |
| 1.2.3 Study Dose Selection | 29 |
| 1.2.4 Risk-Benefit Assessment | 30 |
| 1.2.5 Potential Risks | 31 |
| 1.2.5.1 Anaphylaxis and Serious Allergic Reactions | 32 |
| 1.2.5.2 Injection Site Reactions | 32 |
| 1.2.5.3 Immune Complex Disease | 32 |
| 1.2.5.4 Infections | 33 |
| 1.2.5.5 Malignancy | 33 |
| 1.2.5.6 Hepatic Function Abnormality | 34 |
| 1.2.5.7 Failure of Vaccination | 34 |
| 1.2.5.8 Potential for Drug-Drug Interactions | 34 |
| 1.2.5.9 Potential Risk to Fetal Development | 35 |
| 2 STUDY OBJECTIVES AND ENDPOINTS | 35 |
| 2.1 Phase 1b Multiple Ascending Dose | 36 |
| 2.2 Phase 2 Proof of Concept | 38 |
| 3 STUDY PLAN | 39 |
| 3.1 Study Design | 39 |
| 3.1.1 Multiple Ascending Dose Phase 1b | 40 |
| 3.1.1.1 Dose Escalation for the MAD Portion | |
| 3.1.1.2 Dose Limiting Toxicity (DLT) | |
| 3.1.1.3 DMC Recommendations | 41 |
| 3.1.2 POC Phase 2 | |
| 3.1.2.1 BOS161721 POC Dose Selection and Justifica | tion41 |

| 3.1.2.2 | POC Study Design | 42 |
|---------|-------------------------------------------------------------|----|
| 3.2 | Randomization and Blinding | 42 |
| 3.3 | Study Schematic | 44 |
| 3.4 | Schedule of Assessments | 45 |
| 3.5 | End of Study | 49 |
| 4 PC | OPULATION | 49 |
| 4.1 | Participant Recruitment | 49 |
| 4.2 | Number of Patients | 49 |
| 4.3 | Patient Screening | 49 |
| 4.4 | Inclusion Criteria | 49 |
| 4.5 | Exclusion Criteria | 52 |
| 4.6 | Concomitant Medications | 54 |
| 4.6.1 | Corticosteroid | 54 |
| 4.6.2 | Other Prohibited and/or Restricted Treatments | 55 |
| 4.7 | Women of Childbearing Potential | 56 |
| 4.7.1 | Determination of Menopause | 56 |
| 4.7.2 | Contraception | 56 |
| 4.8 | Deviation from Inclusion/Exclusion Criteria. | 57 |
| 4.8.1 | Patient Withdrawal and Replacement | 57 |
| 5 S | ΓUDY PROCEDURES | 57 |
| 5.1 | Screening. | |
| 5.1.1 | Retesting During Screening Period | 59 |
| 5.2 | Enrollment/Randomization and Day 0 Treatment | 59 |
| 5.3 | Treatment Period/Follow-Up Visits | 60 |
| 5.4 | Safety Follow-Up Visits | 61 |
| 5.5 | Premature Discontinuation. | 61 |
| 6 A | SSESSMENTS | 62 |
| 6.1 | Medical History, Demographic and Other Baseline Information | 62 |
| 6.2 | Safety Assessments | 63 |
| 6.2.1 | Laboratory Assessments | 63 |
| 6.2.1.1 | Pregnancy testing | 64 |
| 6.2.1.2 | 2 Tuberculosis Screening | 65 |
| 6.2.2 | Adverse Events | 65 |
| 6.2.2.1 | Definitions | 65 |
| 6.2.2.2 | Recording of Adverse Events | 66 |
| 6.2.2.3 | Severity of Adverse Events | 66 |
| 6.2.2.4 | Causality of Adverse Events | 66 |
| 6.2.2.5 | Seriousness of Adverse Events | 67 |
| 6.2.2.6 | Adverse Events of Special Interest | 68 |
| 6.2.2.7 | Reporting of Adverse Events | 71 |
| 6.2.2.8 | Follow Up of Adverse Events | 73 |

| Clinical Study Protocol: BO | OS161721-02 |
|-----------------------------|--------------------|

| 6.2.3 | Vital Signs | 73 |
|---------|--------------------------------------------------------------|----|
| 6.2.4 | 12-Lead Electrocardiograms | 73 |
| 6.2.5 | Physical Examinations | 74 |
| 6.2.6 | C-SSRS | 74 |
| 6.2.7 | Injection Site Reactions | 74 |
| 6.2.8 | Immunogenicity | 74 |
| 6.3 | Efficacy Assessments | 75 |
| 6.3.1 | SLEDAI-2K | 75 |
| 6.3.2 | BILAG 2004 | 75 |
| 6.3.3 | PGA of Disease Activity | 75 |
| 6.3.4 | Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response | 76 |
| 6.3.4.1 | SRI-4 Response | 76 |
| 6.3.4.2 | SRI-5 and SRI-6 Response | 76 |
| 6.3.4.3 | BICLA Response | 76 |
| 6.3.5 | CLASI Response | 76 |
| 6.3.6 | ACR-28 Joint Count | 77 |
| 6.4 | Other Variables | 77 |
| 6.4.1 | SLICC/ACR Damage Index | 77 |
| 6.4.2 | PROs | 77 |
| 6.5 | Pharmacokinetic Assessments | 77 |
| 6.6 | Pharmacodynamic Assessments | 77 |
| 6.7 | Pharmacokinetic/Pharmacodynamic Relationship | 78 |
| 6.8 | Protocol Deviations | 78 |
| 7 S7 | ΓUDY DRUG MANAGEMENT | 78 |
| 7.1 | Description | 78 |
| 7.1.1 | Formulation | 78 |
| 7.1.2 | Storage | 78 |
| 7.2 | Packaging and Shipment | 78 |
| 7.3 | Dose and Administration | 78 |
| 7.4 | Accountability | 79 |
| 7.5 | Prohibited Concomitant Therapy | 79 |
| 7.6 | Compliance | 79 |
| 8 S7 | TATISTICS | 79 |
| 8.1 | Sample Size | 80 |
| 8.2 | Statistical Methods | 81 |
| 8.2.1 | Analysis Populations | 81 |
| 8.2.2 | Demographics and Baseline Characteristics | 81 |
| 8.2.3 | Primary Efficacy Endpoint(s) | 81 |
| 8.2.4 | Secondary Efficacy Endpoint(s) | 82 |
| 8.2.5 | Analysis of Safety | 82 |
| 8.2.5.1 | Safety Analysis | 82 |

| Clinical Study Protocol: BO | OS161721-02 |
|-----------------------------|------------------|
| Protocol Date and Version: | 23 July 2019: V6 |

| 8.2.6 | Pharmacokinetic and Pharmacodynamic Data | 82 |
|---|---|---|
| 8.2.6.1 | Analysis of Pharmacokinetic Data | |
| 8.2.6.2 | Analysis of Pharmacodynamic Data | 83 |
| 8.2.6.3 | Population Pharmacokinetic Analysis or PK/PD Modeling | 83 |
| 8.3 Inter | rim Analysis and Power | 83 |
| 9 ETHIC | S AND RESPONSIBILITIES | 83 |
| 9.1 Goo | d Clinical Practice | 83 |
| 9.2 DM | C | 83 |
| 9.3 Insti | tutional Review Board/Independent Ethics Committee | 84 |
| 9.4 Info | rmed Consent | 84 |
| 9.5 Rec | ords Management | 85 |
| 9.6 Sour | ce Documentation | 86 |
| 9.7 Stud | y Files and Record Retention | 86 |
| 10 AUDIT | ING AND MONITORING | 86 |
| 11 AMEN | DMENTS | 86 |
| 12 STUDY | Y REPORT AND PUBLICATIONS | 87 |
| 13 STUDY | Y DISCONTINUATION | 87 |
| 14 CONFI | DENTIALITY | 87 |
| 15 REFER | ENCES | 89 |
| 16 APPEN | IDICES | 93 |
| <b>APPENDIX</b> | 1 NAMES OF STUDY PERSONNEL | 93 |
| <b>APPENDIX</b> | DECLARATION OF HELSINKI | 94 |
| <b>APPENDIX</b> | COMMONLY USED CORTICOSTEROID EQUIVALENTS | 98 |
| <b>APPENDIX</b> | 4 MEDICATION WASHOUT PERIODS | 99 |
| <b>APPENDIX</b> | BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA) | 100 |
| <b>APPENDIX</b> | 16 INJECTION SITE REACTION GRADING SCALE | 101 |
| <b>APPENDIX</b> | 7 OPIOID ORAL MORPHINE MILLIGRAM EQUIVALENTS OF | |
| | IONLY USED OPIOIDS | 102 |
| | SCHEDULE OF ASSESSMENTS - PHASE 1B MULTIPLE | |
| | NDING DOSE | |
| APPENDIX | PROTOCOL SUMMARY OF CHANGES | 110 |
| | LIST OF IN-TEXT TABLES | |
| Table 1. | Schedule of Assessments - Phase 2 Proof of Concept (POC) | 45 |
| Table 2. | Laboratory Tests | 63 |
| Table 3. | Causality Definitions | 67 |
| Table 4 | Schedule of Assessments - Phase 1b - Multiple Ascending Dose | 105 |


# LIST OF IN-TEXT FIGURES

| Figure 1. | Individual pSTAT3 C <sub>min</sub> Levels Versus Dose | 30 |
|-----------|-------------------------------------------------------|----|
| Figure 2. | Study Diagram for MAD Phase 1b and POC Phase 2 | 44 |


# LIST OF ABBREVIATIONS

ACR American College of Rheumatology

ADA anti-drug antibody
ADL activities of daily living

AE adverse event

AIDS acquired immune deficiency syndrome

ALT alanine aminotransferase
ANA antinuclear antibodies
ANC absolute neutrophil count
ANOVA analysis of variance

ANCOVA analysis of covariance APL antiphospholipid

AST aspartate aminotransferase

AUC area under the concentration-time curve

AZA azathioprine

BICLA BILAG-based Composite Lupus Assessment

BILAG British Isles Lupus Assessment Group

BMI body mass index
BP blood pressure
BUN blood urea nitrogen

BW body weight C complement

C-SSRS Columbia Suicide Severity Rating Scale

CD cluster of differentiation

CK creatine kinase

C<sub>L</sub> systematic clearance

CLASI Cutaneous Lupus Erythematosus Area and Severity Index

C<sub>max</sub> maximum plasma concentration

CMH Cochran-Mantel-Haenszel

CS corticosteroids
CSR clinical study report
DILI drug-induced liver injury
DLT dose-limiting toxicity
DMC data monitoring committee

dsDNA double-stranded deoxyribonucleic acid

ECG electrocardiogram
EOT end of treatment

eCRF electronic case report form

F female

CCI


Fc fragment crystallizable

FDA Food and Drug Administration
FSH follicle stimulating hormone

GCP Good Clinical Practice

eGFR estimated glomerular filtration rate

GLP Good Laboratory Practice

GWAS genome-wide association studies

γc gamma chain HBV hepatitis B virus

hCG human chorionic gonadotropin

HCl hydrochloride HCV hepatitis C virus

HIV human immunodeficiency virus

HR heart rate

HRT hormone replacement therapy

IA interim analysis

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonization

IEC Independent Ethics Committee

Ig immunoglobulin

IL interleukin

IL-21R interleukin 21 receptor

IM intramuscular IFNγ interferon gamma

INR International Normalized Ratio
IRB Institutional Review Board

IUD intrauterine device

IV intravenous

IVRS interactive voice response system

JAK Janus kinase kg kilogram

KLH keyhole limpet hemocyanin LOCF last observation carried forward

M male

mAb monoclonal antibody
MAD multiple ascending dose

MAPK mitogen-activated protein kinase

MedDRA Medical Dictionary of Regulatory Activities

MS multiple sclerosis


MTX methotrexate

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NIAID/FAAN National Institute of Allergy and Infectious Diseases/Food Allergy and

Anaphylaxis Network

NK natural killer

NOAEL no observed adverse event level

NO nitric oxide

NSAID nonsteroidal anti-inflammatory drug

OTC over-the-counter
PD pharmacodynamics
PEF peak expiratory flow

PGA Physician's Global Assessment

PK pharmacokinetics
POC proof of concept
PP per protocol

PR (interval) from onset of the p-wave to the end of the r-wave

pSS primary Sjögren's syndrome

pSTAT3 phosphorylated signal transducer and activator of transcription 3

PT preferred term

QRS (interval) from the onset of the q-wave to the end of the s-wave
QT (interval) from onset of the QRS complex to the end of the T wave
QTcF QT interval corrected for heart rate using Fridericia's formula

QFT-G QuantiFERON-TB Gold In-Tube

RA rheumatoid arthritis

RR (interval) from the onset of the r-wave to the onset of the next consecutive r-

wave

SAD single ascending dose SAE serious adverse event SAP statistical analysis plan

SC subcutaneous

SDMT safety data monitoring board

SLE systemic lupus erythematosus SLEDAI-2K SLE Disease Activity Index 2000

SLICC Systemic Lupus International Collaborating Clinics

Sm Smith

SOC system organ class
SRI-4 SLE Responder Index 4
SRI-5 SLE Responder Index 5
SRI-6 SLE Responder Index 6

SS safety analysis set


SSA Sjögren syndrome-A (Ro) SSB Sjögren syndrome-B (La)

STAT3 signal transducer and activator of transcription 3 SUSAR suspected unexpected serious adverse reaction

t<sub>1/2</sub> terminal elimination half-life

TB tuberculosis

TDAR T-cell dependent antibody response

Tfh T-follicular helper

Th T-helper
TK toxicokinetics

T<sub>max</sub> first time to maximum concentration

Treg regulatory T-cell ULN upper limit of normal

US United States

Vd volume of distribution

WBC white blood cell

WHO World Health Organization
WOCBP women of childbearing potential

YTE triple mutation


# 1. INTRODUCTION AND RATIONALE

#### 1.1 Indication

BOS161721 is a humanized monoclonal antibody (mAb), which binds to and inhibits interleukin-21 (IL-21) bioactivity, and is being developed for the treatment of moderately to severely active systemic lupus erythematosus (SLE) in adults.

# **1.2** Background and Rationale

#### 1.2.1 Overview of the Disease State

SLE is a chronic inflammatory autoimmune disease that has variable manifestations in multiple organ systems and follows a relapsing and remitting course. The disease process includes abnormal immune responses mediated by tissue-binding autoantibodies and immune complex deposition, giving rise to tissue damage often resulting in end organ disease and even mortality. Survival of SLE has improved due to earlier detection, improved overall medical care, and standardized SLE treatment with corticosteroids (CS), immunosuppressants, and cytotoxic agents. However, some of the morbidity in patients with SLE is related to its treatment. Comparison of early and late outcomes in patients with SLE demonstrate that death in early disease is most commonly due to infections and active SLE causing multi-system organ damage, while thromboses were the most common cause of death during later disease.<sup>2</sup>

The reported prevalence of SLE in the United States (US) is 20 to 70 cases per 100,000 people.<sup>3</sup> More than 90% of cases of SLE occur in women, frequently starting at childbearing age. Women of color are disproportionately affected by SLE. This suggests multiple genetic and environmental factors are at play. Accordingly, a multifactorial view of the immunopathogenesis of SLE suggests more than 1 area of interest, including breach in central tolerance in the adaptive arm of the immune system, peripheral amplification of the autoimmune response by the innate immune system, and local processes in the target organ that facilitate end-organ disease.<sup>4</sup>

### **1.2.2 BOS161721 Development**

Boston Pharmaceuticals is developing BOS161721 for the treatment of SLE. BOS161721 is a humanized immunoglobulin G1 (IgG1) mAb with extended half-life directed against human IL-21.

Murine mAb 19E3, the progenitor of BOS161721, was generated using mouse hybridoma technology. 19E3 has subpicomolar (pM) affinity to human IL-21 and was selected for its potent neutralization of IL-21 bioactivity. BOS161721 was generated by the humanization of mAb 19E3 where its complementarity-determining regions were grafted onto a human IgG1 kappa backbone. The fragment crystallizable (Fc) portion of BOS161721 contains a YTE (M252Y/S254T/T256E triple mutation) in the constant domain of the IgG1 heavy chain that was introduced into the parental molecule, 19E3, intended to prolong the *in vivo* terminal elimination half-life (t½) of the mAb. Thus, BOS161721 retains sub-pM binding to IL-21 and prevents IL-21 from binding to the IL-21 receptor (IL-21R), inhibiting IL-21 bioactivity.


BOS161721 binds to human IL-21 and Cynomolgus monkey IL-21, which are highly homologous, and neutralizes the bioactivity of both. BOS161721 is specific for IL-21 as it does not bind to or inhibit the other gamma-chain (γc) family of cytokines, and acts to specifically neutralize the IL-21 pathway. In *in vitro* studies, BOS161721 inhibited downstream IL-21-induced signaling, IL-21-induced plasma cell differentiation, and IL-21-induced natural killer (NK) cell activation. In *in vivo* studies, BOS161721 significantly inhibited the T-cell dependent antibody response (TDAR) to immunization with a protein antigen as well as B-cell expansion following a second protein antigen immunization in Cynomolgus monkeys.

#### **1.2.2.1 Interleukin-21**

IL-21 is an inflammatory cytokine, which belongs to a family of cytokines that also includes IL-2, IL-4, IL-7, IL-9, and IL-15, all of which bind to private receptors in complex with the common cytokine receptor yc. 6 Most cytokines in this family are critically important for both the maintenance and function of T-cell and B-cell responses. IL-21 signals through a receptor complex consisting of its own private receptor, the IL-21R and vc.<sup>6,7</sup> Engagement of the IL-21R/γc complex leads to the activation of several signaling pathways, including the Janus kinase/signal transducer and activator of transcription, mitogen-activated protein kinase (MAPK) and phosphoinositide 3-kinase pathways. EL-21 is produced mainly by T-cells and NK T-cells, but neutrophils have also been reported to produce IL-21. 9,10 The IL-21R is expressed on a broad array of cell types, including B-cells, T-cells, NK-cells, macrophages and dendritic cells, as well as other hematopoietic and nonhematopoietic cells such as fibroblasts, keratinocytes, and intestinal epithelial cells.<sup>9,11</sup> Activation of signal transducer and activator of transcription 3 (STAT3) via phosphorylation is critical in regulating human B-cell responses to IL-21<sup>12</sup>; phosphorylated STAT3 (pSTAT3) forms a homodimer, which translocates to the nucleus where it initiates transcription of the IL-21 gene, forming an autocrine loop for IL-21 production via STAT3 phosphorylation. <sup>13</sup> In addition, IL-21 has been shown to upregulate expression of its own receptor <sup>14</sup> and induces an autocrine feedback loop. <sup>15</sup>

IL-21 modulates various aspects of immune function. It promotes cluster of differentiation 4 (CD4+) T-cell differentiation and promotes the generation of T-helper (Th)17<sup>16</sup> and T-follicular helper (Tfh) cells. <sup>15,17</sup> In mice, IL-21 has been shown to regulate the balance between Th17 and regulatory T-cell (Treg), in that it increases Th17, while inhibiting Treg differentiation. <sup>18</sup> Less is understood with regards to human Tregs, although IL-21 has been reported to counteract Treg suppression of human effector T-cells <sup>19</sup> and blockade of IL-21 promotes Treg generation in a murine model of graft versus host disease induced by human T-cells. <sup>20</sup> IL-21 upregulates CD8+ T-cell and NK-cell expansion and cytolytic activity by increasing granzyme B and perforin. <sup>21,22</sup> IL-21 also has been reported to increase granzyme B in plasmacytoid dendritic cells and B-cells resulting in inhibition of T-cell responses. <sup>23,24</sup> IL-21 also has a variety of effects on nonhematopoietic cells, such as stromal cells and induces inflammation through matrix metalloproteinase release by gut intestinal fibroblasts. <sup>25</sup>

One principal non-redundant role of IL-21 is the promotion of B-cell activation, differentiation, or death during humoral immune responses. <sup>14</sup> Furthermore, increased IL-21 production is characteristic of several autoimmune diseases and is likely to contribute to autoantibody production as well as pathologic features of autoimmune disease. <sup>26</sup> The critical role of IL-21 in promoting humoral and other immune responses makes it an important focus of potential


therapeutic interventions in conditions characterized by overproduction of pathogenic autoantibodies. IL-21 production by Tfh cells in humans is believed to play a major role in driving the autoantibody production through its role in plasma cell differentiation. Importantly, Tfh cell populations are expanded in patients with autoimmune diseases such as lupus, bullous pemphigoid, rheumatoid arthritis (RA) and primary Sjögren's syndrome (pSS) and have been reported to correlate with IL-21 levels, autoantibodies, and disease severity. <sup>26,27,28,29</sup> Furthermore, loss of number and functionality of Tregs has been associated with autoimmune diseases such as SLE and giant cell arteritis, which IL-21 is expected to modulate. <sup>30,31</sup> Thus, neutralization of IL-21 in settings of autoimmunity is expected to impact several cell populations believed to be involved in the pathogenesis of autoimmune disorders including SLE.

BOS161721 selectively binds IL-21 with high affinity to neutralize IL-21, and due to its pleiotropic nature, neutralization of IL-21 is expected to impact several cell populations believed to be involved in the pathogenesis of SLE. Importantly, patients with SLE have elevated IL-21 plasma levels that correlate with the severity of the disease. Recently, genome-wide association studies (GWAS) have provided convincing evidence that the chromosomal 4q 27 region harbors the IL-21 genes and is associated with chronic inflammatory disorders, including SLE.<sup>29</sup>

#### 1.2.2.2 Preclinical Studies

The pharmacokinetics (PK) of BOS161721 were characterized following single-dose intravenous (IV) administration of BOS161721 (0.01 to 30 mg/kg) in male Cynomolgus monkeys or repeat, every 2 weeks IV administration (15 to 100 mg/kg) and subcutaneous (SC) administration (50 mg/kg) in male and female Cynomolgus monkeys. Systemic exposure was approximately dose-proportional within the tested dose range. SC bioavailability was determined to be 64.3%.

Two single-dose (IV) non-good laboratory practice (GLP) studies conducted in Cynomolgus monkeys evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), and immunogenicity of BOS161721. Following a single IV administration (slow bolus), there were no BOS161721-related adverse changes, resulting in a no-observed-adverse-effect-level (NOAEL) value of 30 mg/kg, the highest dose tested among 2 studies.

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) administration for 3 months (a total of 7 doses).




An additional GLP, repeat-dose toxicity study was conducted in Cynomolgus monkeys (4 males and 4 females per dose group) following every 2 weeks (Q2W) administration by SC (10, 30, and 100 mg/kg) injection for a total of 14 doses.

There were no BOS161721-related effects on survival, clinical signs, male body weights, ophthalmologic parameters, electrocardiogram (ECG) findings, clinical pathology, macroscopic observations, organ weights, or microscopic observations.

#### 1.2.2.3 Clinical Studies

BOS161721-01 was a double-blind, Phase 1, single ascending dose (SAD) study to assess the safety, PK, and PD of BOS161721 in healthy subjects. The primary objective of the study was to characterize the safety and tolerability of IV and SC SADs of BOS161721 in an otherwise healthy subject population without concomitant illnesses, immune abnormalities, or concomitant medications. Secondary objectives included characterization of the PK and immunogenicity of BOS161721, and exploratory objectives included the evaluation of the effect of BOS161721 on TDAR to keyhole limpet hemocyanin (KLH) (primary and secondary immunizations) in healthy subjects, the effects of BOS161721 on plasma levels of IL-21 (free and bound), and the evaluation of the effect of BOS161721 on IL-21 gene expression (via gene signature) in blood. This study consisted of 8 cohorts. Subjects were randomized in a 3:1 ratio (BOS161721: placebo) and received either a single dose of BOS161721 (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) or placebo, with safety follow-up. For the first cohort, after the first 2 subjects were dosed (1 active and 1 placebo), there was a minimum gap of 48 hours before the remaining subjects from that cohort were dosed, to allow for an initial review of any emerging safety and tolerability data. For all cohorts, escalation to the next dose was not sooner


than 8 days after all the subjects in the prior cohort had been dosed and were based on a review of at least 7 days of safety and tolerability data by the Safety Data Monitoring Team (SDMT).

Blood samples were collected at every in-house study visit for BOS161721 concentration determinations. Blood samples were also collected for determination of IL-21 plasma levels (free and total). Safety was assessed based on the occurrence of treatment-emergent AEs, hepatic function abnormality, and acute and delayed hypersensitivity reactions. Other safety variables included ECGs, vital signs (blood pressure [BP], heart rate, and temperature), safety laboratory assessments, blood sampling for ADAs, total IgG and immunoglobulin M (IgM) levels, CD4+ count, and full and targeted physical examinations. Overall, there were no clinically significant findings from this study. Adverse events reported as related to the study drug, particularly infections, were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. There was 1 serious adverse event (SAE; death due to pulmonary embolism) that occurred 127 days after a single administration of 240 mg SC dose of BOS161721. The causality of this single SAE was not attributed to study drug and further information can be found in the Investigator's Brochure. Final PK data from the SAD study demonstrates BOS161721 has a mean t½ ranging from 80 to 87 days for doses of ≥ 30 mg in healthy subjects.

# 1.2.3 Study Dose Selection

Doses have been selected for the multiple ascending dose (MAD) Phase 1b portion based on a 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01); the SDMT reviewed the blinded safety data from subjects for each dose cohort (8 cohorts, evaluating 1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg), along with the accumulated safety and available PK/PD data from all subjects in the previous dose cohorts, to make a decision on whether to proceed to the next higher dose level, repeat a dose level, or stop dose escalation. Overall, there were no clinically significant safety or tolerability findings from this study.

Based on the Day-90 interim cut of the PK and biomarker data in the BOS161721-01 study, the recommended doses for evaluation in the MAD portion of this study are 20, 60, and 120 mg SC monthly. This dose recommendation is supported by evidence of linear PK with BOS161721 resulting in a median first time to maximum concentration (T<sub>max</sub>) of 6 days and an apparent terminal half-life of 44 days. Furthermore, pSTAT3 suppression, a marker of IL-21 target engagement, follows a similar time course of the mAb levels, with maximal and sustained suppression apparent with doses greater than 30 mg SC (Figure 1).


pSTAT3 cmin (percent pSTAT3+ lymphocytes, stimulated) 60 pSTAT3 cmin Route IV ▲ SC 20 100 0 50 150 200 250 Dose (mg)

Figure 1. Individual pSTAT3 C<sub>min</sub> Levels Versus Dose

IV = intravenous, pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SC = subcutaneous

All doses selected for the MAD portion are projected not to exceed the mean exposure of that achieved following the highest single dose of 240 mg SC administered in the Phase 1 SAD study. Cohort 1 will include randomized treatment to the 20 mg dose. Based on the staggered study design, the data monitoring committee (DMC) will perform a scheduled review of safety data and sequentially consider dose escalation for Cohorts 2 and 3. In addition, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the proof of concept (POC) Phase 2 portion. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD portion (see Section 3.1.2.1 for the chosen POC dose and justification).

#### 1.2.4 Risk-Benefit Assessment

The available preclinical data on BOS161721, the findings in clinical study BOS161721-01, and existing clinical information on IL-21 inhibitors suggest that the present clinical study has an acceptable risk-benefit ratio. In this study, the risk-benefit assessment of BOS161721 in adult patients with moderately to severely active SLE will be ongoing, with step-wise evaluations during the staggered MAD portion. The DMC used in this study is charged with assessing such actions in light of an acceptable benefit-risk profile for BOS161721 as an anti-IL-21 mAb.


Formal DMC monitoring meetings will occur as described in the DMC Charter. Two weeks after Cohort 1 has received a second dose of study drug, the DMC will evaluate the safety and tolerability data from Cohort 1 to determine the recommended dose for Cohort 2. Two weeks after 8 patients in Cohort 2 receive a second dose, the DMC will determine if dose escalation to Cohort 3 can proceed. Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 during the MAD part of study. Thereafter, DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter. With the agreement of the DMC and sponsor, this schedule may be modified depending on the rate of patient accrual. Additional details can be found in the DMC Charter.

The benefit of participation for all patients in this study is close monitoring of their medical condition and safety of their treatment. Those randomized to the active treatment arm may potentially experience improvement in their SLE disease. Those randomized to the placebo (in combination with standard of care) arm are not expected to obtain any additional benefit, beyond those of their background treatment, though close monitoring of their medical condition and safety may itself be associated with improving their SLE.

#### 1.2.5 Potential Risks

Potential risks based on the mechanism of action of BOS161721 include infections, risks associated with the administration of any foreign protein or biologic agent, including injection site reaction, anaphylaxis, serious allergic reaction, and development of ADAs. ADAs could result in immune complex disease (with manifestations such as arthralgias, serum-sickness, and vasculitis), or altered BOS161721 levels or activity. Further details can be found in the current Investigator's Brochure (IB) for BOS161721, which contains comprehensive toxicology, preclinical and clinical information on BOS161721.

Two investigational drug products are considered to be in the same pharmacological class as BOS161721 based on interruption of signaling through the IL-21 signaling pathway. No potential risk generalizable across the class has been observed with these investigational products. Based on the clinical Phase 1 SAD study (BOS161721-01), AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc.), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs.

The majority of IgG elimination occurs via intracellular catabolism, following fluid-phase or receptor-mediated endocytosis. This type of endocytosis and elimination is a form of target-mediated disposition where the interaction of the drug and its pharmacological target (eg, a target receptor) serves as a significant contributor to the kinetics of antibody distribution and elimination. Renal elimination, which is a primary pathway of clearance of small-molecule drugs, is relatively unimportant for IgG, as its large size prevents efficient filtration through the glomerulus. Secretion into the bile is an important pathway of elimination of IgA antibodies, but this route is not a significant contributor to the elimination of IgG antibodies. Thus, risk to renal and hepatic systems due to metabolism of BOS161721 is low.<sup>33</sup>


# 1.2.5.1 Anaphylaxis and Serious Allergic Reactions

As with the administration of any foreign protein and/or other biological agents, acute hypersensitivity reactions, including acute anaphylactic/hypersensitivity, severe allergic, and anaphylactoid reactions may follow infusion of mAbs and can be caused by various mechanisms. These acute hypersensitivity reactions may be severe and result in death.

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria,<sup>34</sup> and are discussed in Section 6.2.2.6.1.

Based on the Phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed.

Patients with a known history of allergy or severe hypersensitivity reaction to any component of BOS161721 formulation or patients with a history of anaphylaxis to any other biological therapy such as mAbs will be excluded from studies with BOS161721. In addition, appropriate drugs and medical equipment to treat acute hypotensive, bronchoconstrictive, or anaphylactic reactions will be immediately available at the unit and study personnel will be trained to recognize and treat these reactions.

# 1.2.5.2 Injection Site Reactions

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC for 3 months (a total of 7 doses). There were no injection site reactions in animals dosed subcutaneously. Further, there were no reports of injection site reactions in the 26-week GLP toxicology study in Cynomolgus monkeys.

Based on the Phase 1 SAD study (BOS161721-01), incidence of injection site reactions in subjects who received BOS161721 was similar to placebo.

Patients will be monitored for local injection site reactions in this study. See Section 6.2.7.

# 1.2.5.3 Immune Complex Disease

The potential risk of immune complex disease for BOS161721 is theoretical, based on the known risks associated with mAbs. The administration of a mAb can result in the formation of ADAs. Administration of the mAb in the presence of ADA may result in the formation of circulating antibody-antigen complexes potentially resulting in altered BOS161721 levels or activity or deposition of the complexes in microvasculature. Complement is frequently involved in the latter setting, and the breakdown products of complement attract polymorphonuclear leukocytes to the site of deposition where they can provoke local tissue damage through specific or nonspecific release of enzymes. Two of the more common end-organ targets are the blood vessels (vasculitis) and kidney (nephritis). These clinical manifestations represent immune complex disease or Type III hypersensitivity. Although BOS161721 is a humanized mAb, ADAs may develop; however, the likelihood of occurrence of immune complex disease with BOS161721 is low. The findings of immune complex disease are typically reversible when mAb administration stops and the antibody-antigen complexes are cleared from the body.


Based on the Phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed.

#### 1.2.5.4 Infections

BOS161721 is expected to diminish the activity of T-cell, B-cell and NK-cell lines. Like other medications modulating immune response, BOS161721 may increase the potential risk for infection, including serious infections. IL-21 produced by CD4+ Th cells is required to sustain the anti-viral function of CD8+ T-cells against chronic viral infections. Nonclinical evidence suggests that the risk of chronic viral infection recurrence or increased severity may occur with IL-21 inhibition.<sup>35</sup>

These conditions will be fully characterized with clinical descriptions and routine laboratory and/or specialty testing and treated where indicated with appropriate local standard of care.

Patients with a history of opportunistic infection, including recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years, or any other underlying pathology predisposing to serious infection, are excluded from studies with BOS161721 (for further details please refer to the current IB for BOS161721).

Patients will be assessed for hepatitis B, and C, and HIV-1/2 combination, at screening.

# Cryptosporidium Infection

Cryptosporidium infection was noted in patients with an IL-21 receptor loss-of-function gene mutation and similar findings of cryptosporidium infection have been observed in immunosuppressed liver transplant and human immunodeficiency virus patients. Since BOS161721 is expected to diminish the immunosurveillance activity of T-cell, B-cell, and NK-cell lines, a similar risk is biologically plausible with prolonged exposure to BOS161721.

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells,  $^{37}$  patients with a CD4+ count < 500 cell/mm $^3$  were excluded from the Phase 1 SAD study (BOS161721-01), and CD4 + < 350 cells/mm $^3$  will be excluded from the MAD/POC parts of the study. Patients exposed to investigational product who develop diarrhea during the course of the study should immediately undergo an assessment for opportunistic infection including stool for ova and parasites and stool examination for cryptosporidium. Positive cryptosporidium in stool sample at screening is an exclusion. Treatment by the investigator where indicated should be guided by findings and be consistent with local standard of care.

Based on the Phase 1 SAD study (BOS161721-01), infections in subjects who received BOS161721 was not observed.

### 1.2.5.5 Malignancy

The stimulatory effect of IL-21 on NK cells and CD8+ T-cells suggests the cytokine may have anti-tumor activity. Nonclinical studies have demonstrated significant anti-tumor effects of IL-21 in a number of tumor models. IL-21 therapy of human metastatic melanoma and renal cell carcinoma has demonstrated POC with significant increases in levels of perforin, granzyme B,


and interferon gamma (IFNγ) expression in CD8+ T-cells and NK T-cells. Clinical response has been limited in these generally unmanageable diseases.

The impact of treatment with anti-IL-21 therapy on the development or growth of malignancies is not known; however, as with other immunomodulatory biologic agents, treatment with BOS161721 may result in an increase in the risk of malignancies. NK cell suppression by IL-21 neutralization may represent a biological mechanism for a potential risk for malignancy. Patients with a history or current diagnosis of cancer within the past 5 years, with the exception of non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy, are excluded from the study.

Based on the Phase 1 SAD study (BOS161721-01), malignancy in subjects who received BOS161721 was not observed.

### 1.2.5.6 Hepatic Function Abnormality

There is no substantial evidence suggesting BOS161721 is associated with liver function abnormality. However, as a precaution, patients with a history of abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST >  $2 \times \text{upper limit of normal [ULN]}$ ; total bilirubin >  $1.5 \times \text{[ULN]}$  and judged by the investigator to be clinically significant) were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from this trial. Patients with a positive hepatitis B or C test or a history of alcohol dependence will also be excluded.

Based on the Phase 1 SAD study (BOS161721-01), hepatic function abnormality in subjects who received BOS161721 was not observed.

#### **1.2.5.7** Failure of Vaccination

IL-21 is a key cytokine in development of B-cells into immunoglobulin-secreting plasma cells. Abnormal signaling through the IL-21R/Janus Kinase (JAK)3/signal transducer and activator of transcription (STAT3) pathway leads to defective humoral immune responses to both T-dependent and T-independent antigens and impairs the establishment of long-lasting B-cell memory. Abnormal signaling through the pathway has been related to decreased specific antibody responses following vaccination, and to increased susceptibility to encapsulated bacterial infections.<sup>38</sup>

The effect of BOS161721 was evaluated in *in vivo* single dose studies in Cynomolgus monkey in which the animals received vaccination to T-cell dependent KLH antigen to stimulate a TDAR. These *in vivo* studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen in a dose-dependent fashion; however, BOS161721 administration did not affect anti-tetanus toxoid antibody data for IgM, IgG, IgG1, or immunoglobulin E (IgE) during the dosing phase in the same study.

### 1.2.5.8 Potential for Drug-Drug Interactions

Drug-drug interactions were not evaluated in the Phase 1 SAD study (BOS161721-01), which included only healthy adult subjects. Use of prescription medications (with the exceptions of


oral contraceptives), and over-the-counter (OTC) treatments including herbal supplements such as St John's Wort (except multivitamins), in the 2 weeks prior to screening was prohibited in the SAD study.

See Section 4.5 for other specific exclusion criteria which support lowered risk of interactions, and Section 4.6.1 for corticosteroid (CS) dosing. In addition, Section 1.2.5.6 describes considerations for hepatic function for this study.

# 1.2.5.9 Potential Risk to Fetal Development

No data on preclinical reproductive toxicity are available at the time of this study.

# 2 STUDY OBJECTIVES AND ENDPOINTS

This trial has separate objectives and endpoints for the MAD Phase 1b and POC Phase 2 portions of the study. The primary, secondary, and exploratory objectives for each phase, as applicable, are described below with their corresponding endpoints.


# 2.1 Phase 1b Multiple Ascending Dose

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose. | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of AEs and SAEs, related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness</li> <li>Injection site reactions</li> <li>Columbia Suicide Severity Rating Scale (C-SSRS)</li> <li>12-lead ECGs parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> <li>Clinical laboratory results and change from baseline</li> <li>Physical examinations changes from baseline</li> <li>ADAs</li> <li>Study drug exposure/compliance</li> </ul> |
| Secondary | |
| To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PD effects in patients with moderately to severely active SLE. | <ul> <li>Pharmacokinetic Endpoints</li> <li>BOS161721 concentration by visit and time point</li> <li>Maximum observed concentration (C<sub>max</sub>), T<sub>max</sub>, area under the concentration-time curve (AUC), terminal elimination half-life (t<sub>½</sub>), systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>)</li> <li>Pharmacodynamic Endpoints</li> <li>Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype</li> <li>Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit</li> <li>Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit</li> </ul> |





Clinical Study Protocol: BOS161721-02

2.2 Phase 2 Proof of Concept

| OBJECTIVES | | ENDPOINTS |
|---|---|---|
| | Primary | |
| Pr<br>• | | Primary Efficacy Endpoint The proportion of patients with a SRI-4 response at Day 210 (see Section 6.3.4.1) Secondary Efficacy Endpoints The proportion of patients with: SRI-4 response at each visit SRI-5 and SRI-6 response at each visit SRI-5 and SRI-6 response at each visit Section 6.3.4.2) a sustained reduction from baseline of oral corticosteroid (CS) (≤ 7.5 mg/day and < Day 0 dose) between Day 150 and Day 210 new or recurrent BILAG flares (≥ 1 qualifying BILAG A or > 1 qualifying BILAG B) through Day 210 PGA worsening a BICLA response a CLASI response medication failures Results and changes from baseline in: CLASI Total number of swollen joints, tender joints, and active joints (swelling and tenderness in the same joint) in the ACR-28 joint count SLEDAI-2K SLICC/ACR damage index Time to medication failure Group mean percent reduction in CS administration from baseline Day 0 dose through Day 210 in patients receiving ≥ 7.5 mg/day prednisone equivalent at Day 0 Duration of longest SRI-4 response Time to first SRI-4 response Time to first SRI-4 response |
| | | Duration of longest SRI-4 response |
| C | 6.4 | • Time to first BILAG flare (≥ 1 new or recurrent BILAG A |
| Sa | Safety | |
| • | To assess safety and tolerability of repeat doses of BOS161721 at the chosen dose administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness</li> <li>Injection site reactions</li> <li>C-SSRS</li> <li>12-lead ECGs parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> </ul> |






### 3 STUDY PLAN

## 3.1 Study Design

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, eligible patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly.

The trial will consist of 2 double-blinded portions: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

SLE disease activity assessment data will be centrally reviewed by medical monitor and sponsor to ensure the scores are clinically meaningful and compliant with specific definition. The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease activity. Further details on the content and methods of data reports by the medical


monitor and sponsor will be outlined in the Medical Data Review Plan along with the processes and procedures that will be followed.

# 3.1.1 Multiple Ascending Dose Phase 1b

The MAD portion will consist of 3 cohorts:

- Cohort 1 (20 mg SC) will include 6 patients
  - o 5 patients will receive BOS161721 (active group) and 1 patient will receive placebo (placebo group)
- Cohorts 2 (60 mg SC) and 3 (120 mg SC) will include 12 patients each
  - o 9 patients in the active group and 3 in the placebo group

Doses selected for each of the 3 cohorts is based on a 90-day safety, tolerability, PK and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. All doses selected for the MAD part of the study are projected not to exceed the mean exposure of that achieved in the SAD study.

#### 3.1.1.1 Dose Escalation for the MAD Portion

The MAD portion of the study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after the DMC evaluation of the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after the DMC evaluation of the safety and tolerability data from Cohorts 1 and 2. Each cohort will continue at their assigned dose level through their respective 6-month treatment periods (See Study Schematic, Section 3.1). If patients discontinue the study in a cohort prior to adequate safety follow-up, he/she may be replaced.

Criteria for dose escalation are further described in the DMC Charter. See Section 3.1.1.2 for additional details about DLTs.

#### 3.1.1.2 Dose Limiting Toxicity (DLT)

Severity of adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs occurring after study drug administration, which are attributable to the study drug, will be considered DLTs:

#### **Hematologic:**

- Grade 4 neutropenia
- Grade 3 neutropenic infection


- Grade 3 thrombocytopenia with bleeding
- Grade 4 thrombocytopenia

# **Non-Hematologic:**

- Grade 3 or above toxicities, persisting after optimal treatment with standard medical therapy (eg, anti-emetics, anti-diarrheals)
- Drug-induced liver injury ([DILI], Hy's Law), as defined in Section 6.2.2.6.3

Investigators should always manage their patients according to their medical judgment which may include interruption of study drug based on the particular clinical circumstances.

#### 3.1.1.3 DMC Recommendations

During scheduled meetings, the DMC will review relevant study data for safety or benefit-risk concern. During the MAD part of the study, the DMC may provide the following recommendations to the sponsor:

- Expanding a cohort at a specific dosing level, or repeating a lower dose in a subsequent cohort
- Continuing a dose level for a given cohort
- Escalating a dose level for a subsequent cohort
- Termination of current or previous cohort(s)

Further dosing in a given cohort will be halted if 2 or more DLTs are identified intra- and inter-patients dosed. For the POC portion, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC Phase 2 part of the study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD portion. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available 30 days after the last patient from Cohort 3 receives the third dose. Details are provided in the DMC Charter.

#### **3.1.2 POC Phase 2**

# 3.1.2.1 BOS161721 POC Dose Selection and Justification

The dose for the POC portion of the study is 120 mg administered SC monthly (a total of 7 doses). The rationale for the BOS161721-02 Phase 2 POC dose selection was based on cumulative safety, tolerability, immunogenicity, PK, and PD data available from an interim analysis (IA) performed during the MAD Phase 1b portion of the trial.


The data cut-off for this IA occurred on CCl and and included all 6 patients and 7 doses from Cohort 1 (20 mg), 12 patients and 6 doses from Cohort 2 (60 mg), and 12 patients and 4 doses from Cohort 3 (120 mg).

The safety analysis focused on incidence and severity of all AEs, SAEs, and pre-determined adverse events of special interest (see Section 6.2.2.6). The DMC and designated unblinded Boston Pharmaceuticals team met on CCI and did not identify any untoward safety signals at any BOS161721 dose levels.

Because there were no safety, tolerability, or immunogenicity trends observed at the time of the IA, the Phase 2 POC dose selection was made based on available PK and PD data. pSTAT3 levels were assessed as the primary PD biomarker of IL-21R signaling levels. This is because IL-21R signaling, upon IL-21 binding, initially involves phosphorylation of JAK1/JAK3 which dissociate from the receptor complex, and phosphorylate STAT3 which translocates to the nucleus and drives IL-21-regulated gene expression.

The 120 mg dose was communicated to site investigators participating in the POC Phase 2 portion, and to Institutional Review Boards (IRBs) and the Independent Ethics Committee (IEC).

# 3.1.2.2 POC Study Design

For the POC part of the study, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio.

As in the MAD part of the study, each patient in the POC portion may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Table 1 and Table 4).

DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.

# 3.2 Randomization and Blinding

This is a randomized, double-blind study.

Patients meeting all inclusion and exclusion criteria will be centrally randomized to either placebo or BOS161721 using an IWRS according to a randomization list generated by an independent, non-study statistician. Randomization will be performed separately for each study portion and separately for each cohort in the Phase 1b and 2 portions as follows:


| Phase/Cohort | Number of Patients | Randomization Ratio BOS161721:Placebo |
|---|---|---|
| Phase 1b/Cohort 1 | 6 | 5:1 |
| Phase 1b/Cohort 2 | 12 | 3:1 |
| Phase 1b/Cohort 3 | 12 | 3:1 |
| Phase 2 | 156* | 2:1 |

<sup>\*</sup>Additional patients may be enrolled to ensure sufficient numbers of patients are in the full analysis set (FAS).

Eligible patients will be assigned to the study portion which is active at time of enrollment. Similarly, patients in the Phase 1b MAD will be assigned to the cohort which is active. Each patient will be assigned a unique randomization number which will not be reused.

All patients, investigators, and study team participants will be blinded to treatment assignment. An independent biostatistician not otherwise involved on the study will be unblinded and prepare materials for the IA, ad hoc analyses as needed, and the DMC safety reviews. The DMC will review unblinded data during safety reviews and the IA. A limited team at Boston Pharmaceuticals will review unblinded results from the Phase 1b MAD portion during the IA to determine the dose that will be used for the Phase 2 POC portion of the study. Details regarding maintenance of the blinding and content of data reviews will be described in the DMC charter or related study documentation.


# 3.3 Study Schematic

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2



A = active drug (BOS161721); P = placebo


# 3.4 Schedule of Assessments

 Table 1.
 Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | Treatment Period Follow-up | | | | | | Safe | ty Follo | w-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| GENERAL ASSESSMENTS | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| SLICC Criteria for SLE | X | | | | | | | | | | | | | |
| Concomitant medication <sup>c</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>d</sup> | | X | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | X | X | X | X | X | X | | | | | |
| SAFETY ASSESSMENTS | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | |
| Chest x-ray <sup>e</sup> | X | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>f</sup> | X | X | | X | | X | | | | | | | | X |
| Injection site reaction assessment | | Xg | | X | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>h</sup> | X | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESSMENTS | | | | | | | | • | | | • | • | | |
| BILAG-2004 Index | X | X | | X | X | X | X | X | X | | | X | X | X |
| SLEDAI-2K | X | Xi | | X | X | X | X | X | X | | | X | X | X |
| PGA | X | X | | X | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | X | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | X | X | X | X | X | X | | | X | X | X |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |


 Table 1.
 Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | T | reatmen | t Period | Follow-u | p | | | Safe | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | - | 10 | 11 | 12 |
| SLICC/ACR Damage Index | | X | | | | | | | X | | | | | |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |
| LABORATORY ASSESSMENT | | | | | | | | | | | | | | |
| CD4+ count | X | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments (hematology and clinical chemistry) <sup>i</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Coomb's test direct <sup>k</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | X | X | | X | | | X | | | | | |
| Plasma CCI | X | X | | X | X | X | X | X | X | | | X | X | X |
| Plasma CCI & CCI | | X | X | X | | X | | | X | | | | | |
| ADA <sup>1</sup> | | X | X | X | X | X | | | X | | | | | X |
| nAb <sup>m</sup> | | | | | | X | | | X | | | | | |
| CCI | | X | X | | | X | | | X | | | | | X |
| CCI | | X | | | | | | | | | | | | |
| CCI | X | X | | X | X | X | X | X | X | | | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> |
| CRP | X | | | | | X | | | | | | | | X |
| Serum pregnancy test (women) | X | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>o</sup> | | X | | X | X | X | X | X | X | | | | | X |
| TB test (QuantiFERON-TB Gold In-Tube) <sup>e</sup> | X | | | | | | | | | | | | | |
| Serology (hepatitis B and C,<br>HIV-1/2 combination) | X | | | | | | | | | | | | | |
| Stool sample <sup>p</sup> | X | | | | | | | | | | | | | |


Table 1. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | T | reatmen | t Period | Follow-u | p | | | Safe | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | to -1 | 0 | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | - | 10 | 11 | 12 |
| Spot urine for protein/creatinine | | | | | | | | | | | | | | |
| ratio | X | X | | X | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | X | X | X | X | X | X | | | X | X | X |
| PK Labs <sup>b</sup> | | | | | | | | | | | | | | |
| Predose | | X | | X | X | X | X | X | X | | | | | |
| Postdose | | | X | | | | | | | X | X | X | X | X |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CC ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; d = day; ECG = electrocardiogram; FSH = follicle stimulating hormone; h = hour; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; m = minute; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; SAE = serious adverse event; SC = subcutaneous; CC ; SLEDAI-2K = SLE Disease Activity

Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; CCl TDAR = T-cell dependent antigen response.

TB = tuberculosis:

<sup>a</sup> Screening assessments will be performed over more than 1 visit.

- PK samples will only be collected at the investigational sites that participate in the PK portion of the study. On PK only days (ie, Day 187 and Day 195 when no laboratory assessments are scheduled) samples will be collected at the investigational sites of the selected countries that participate in the PK portion of the study. Patients not participating in PK are not required to return for investigation site visits on Days 187 and 195.
- <sup>c</sup> Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the dose must be stable for at least 6 weeks prior to Day 0 (randomization day). See Section 4.6.1 for further details.
- Randomization should occur after patient eligibility has been confirmed. The actual randomization procedure can be completed on Day -1 after eligibility confirmation or the morning of Day 0 prior to dosing for logistical purposes.
- <sup>e</sup> If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed at 2 hours postdose.
- <sup>h</sup> Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 187 and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

<sup>i</sup> SLEDAI-2K should be done before randomization and dosing on Day 0 as SLEDAI-2K < 6 is exclusionary.


Table 1. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | Treatment Period Follow-up | | | | | Safe | ty Follo | w-Up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (±3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |

- <sup>j</sup> Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.
- k When clinically indicated for hemolytic anemia.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed (analyzed) if the patient had a positive ADA on Day 90.
- m Ab is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90.
- <sup>n</sup> CCl will not be analyzed during safety follow-up visits.
- <sup>o</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- <sup>p</sup> Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.


# 3.5 End of Study

End of Study (Individual Patient): A patient is considered at the end of study if he/she has withdrawn, prematurely discontinued, or completed all of the study procedures including the last visit.

End of Study (End of trial): The end of the study is defined as the date of the last visit of the last patient in the study globally, or the date of which the last patient withdraws or discontinues if all prior enrolled patients have already completed/withdrawn.

## 4 POPULATION

## 4.1 Participant Recruitment

Advertisements approved by the IRB, and investigator databases, may be used as recruitment procedures for adult men and women with moderately to severely active SLE.

### 4.2 Number of Patients

Approximately 186 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD Phase 1b portion, and approximately 156 additional patients will be randomized in the POC Phase 2 portion. Note that approximately 24 dropouts are assumed.

# 4.3 Patient Screening

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Table 1 and Table 4]) for this study must be performed between Day -28 and Day -1.

#### 4.4 Inclusion Criteria

Patients who meet the following criteria will be considered eligible to participate in this clinical study:

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1


immunologic criterion or Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously

- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
- 5. At screening, the total SLEDAI-2K score must be  $\geq 8$ , including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

- 6. A clinical SLEDAI-2K score of  $\geq$  6 at screening at Day 0. Clinical SLEDAI-2K score is defined as follows:
  - a. Contains points from arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, or vasculitis
  - b. Excludes parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

- 7. Patients must have at least 1 qualifying A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system. If a BILAG B score is due to BILAG number 6, mild skin eruption, the CLASI activity score including erythema and scale/hypertrophy must be  $\geq 3$  excluding points from mucosal ulcers and alopecia.
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - i. "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis defined by BOTH swelling and tenderness in ≥ 6 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living (ADLs) that has been present on several days (> 4 days) cumulatively over the past 30 days, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
      - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):


- Ambulation, toileting, grooming- including bathing and dressing; feeding oneself
- ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis defined by BOTH swelling and tenderness in ≥ 3 joints, (observed or through patient history), with some loss of functional range of movements manifested by effects on instrumental ADLs such as:
  - Cooking, driving, using the telephone or computer, shopping, cleaning, etc., and has been present on several days over the last 30 days, and is present at the time of the screening visit

Note: Hips, shoulders, back, neck, and temporomandibular joints do not count towards the total number of joints with active synovitis.

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in at least 1 other body system for a total of 2 "B" BILAG body system scores.

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to Day 0) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. If AZA, myocophenolate mofetil, mycophenolic acid, hydroxychloroquine, or MTX were discontinued prior to screening, the washout period must be ≥ 12 weeks.
  - c. Corticosteroids (prednisone or prednisone-equivalent) at a stable dose of up to 30 mg/day for at least 6 weeks prior to Day 0 (see APPENDIX 3)
    - i. For patients whose only SLE treatment is CS, the stable CS dose must be ≥ 10 mg/day for at least 6 weeks prior to Day 0 and no more than 30 mg/day at the time of randomization.
    - ii. Topical steroids may be used, but the dose must be stable for at least 6 weeks prior to Day 0. PRN topical steroids are not permitted.
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding


c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks

- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

#### 4.5 Exclusion Criteria

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic sclerosis, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed.
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator or the sponsor or their designee, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study. (See Section 4.6 for prohibited concomitant medication)


- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count < 150/μL at screening
- 16. Platelets < 50,000/mm<sup>3</sup> (50  $\times$  10<sup>9</sup>/L) or < 35,000/ mm<sup>3</sup> (35  $\times$  10<sup>9</sup>/L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation<sup>39</sup>:

GFR = ([1 for male] or [0.85 for female]) 
$$\times$$
 (140 – Age)  $\times$  BW / (72  $\times$  Creatinine)

- 20. Serum ALT and/or serum AST  $> 2 \times$  ULN at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK)  $> 3.0 \times$  ULN at screening, unless it is related to lupus myositis
- 22. Total bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator or the sponsor or sponsor's designee, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (eg, IgG protein) or molecules made of components of monoclonal antibodies
- 25. History substance and/or alcohol abuse or dependence within the past 1 year, at the investigator's judgment
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision)


27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, sponsor or sponsor's designee, would make the patient inappropriate for entry into this study

- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4 or 5 on the C-SSRS
- 31. Current or pending incarceration
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness
- 33. Currently taking a total daily dose of > 30 mg morphine or morphine equivalent (see APPENDIX 7)
- 34. Body mass index (BMI)  $\geq$  40.0

### 4.6 Concomitant Medications

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Patients should stay on stable regimen (not PRN) of other concomitant medications for the treatment of SLE (eg, analgesics, nonsteroidal anti-inflammatory drugs [NSAIDs], statins, ACE inhibitors/ARBs and other antihypertensive drugs), unless changes in these treatments are clinically indicated. Patients should refrain from Tylenol, NSAIDs, and any pain medications including tramadol and other opiates for at least 12 hours before each visit, with the exception of the Screening Visit.

Use of any other drugs for non-SLE conditions, including over-the-counter medications and herbal preparations, should remain stable unless change or addition is clinically necessary. Discussion with the medical monitor prior to initiation of new medication is strongly recommended. Any concomitant therapies must be recorded on the eCRF. Prior and concomitant medication use will be recorded for the 30 days prior to screening until the last follow-up visit. In addition, historical treatment for SLE (including immunosuppressant, anti-malarial, corticosteroid, and/or biologic agent including investigational agents) will be recorded for the 48 weeks prior to screening in the eCRF.

#### 4.6.1 Corticosteroid

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.


A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study. For patients whose only SLE treatment is steroids, their stable steroid dose must be at least 10 mg/day and no more than 30 mg/day for a minimum of 6 weeks at time of randomization on Day 0.

Topical steroids may be used, but the dose must be stable for at least 6 weeks prior to Day 0, and be maintained at a constant dose throughout the study duration until the rashes resolve. PRN topical steroids are not permitted.

Once the patient has received the first dose of study drug (Day 0), tapering of oral steroids will be highly encouraged and should be continually evaluated during the protocol-allowed tapering windows (Day 0 through Day 150) with the target of achieving a CS daily dose of < 7.5 mg and < Day 0 dose between Day 150 and Day 210.

Between Day 150 and Day 210 (ie, within 60 days of primary endpoint assessments), oral CS doses must be held constant.

#### CS Burst for SLE-related Indications

After Day 0 (first dose of study drug), a maximum of 1 oral CS "burst" equivalent to ≤ 40 mg/day prednisone for increased SLE disease activity will be allowed between Day 0 and Day 120, which must be tapered down to the baseline (Day 0) CS dose or lower within 14 days of initiation of the "burst." Any "burst" continuing after Day 120 or occurring after Day 120 is considered a protocol deviation.

• Alternatively, a single intramuscular (IM) dose of methylprednisolone (< 40 mg) is permitted during this period.

#### CS Burst for Non-SLE-related Indications

A single treatment of oral prednisone equivalent of  $\leq 40$  mg/day for 14 days is permitted for a non-SLE indication, though it must be completed prior to Day 120. No long acting steroid injections are permitted.

Note: Treatment with inhaled CS are allowed for the treatment of non-SLE-related indications only (eg, for asthma).

Any other increase from baseline of CS dose or systemic use of CS of any kind (including intra-articular and intravenous administration) are not permitted from Day 0 through Day 210 and will result in the patient being considered a treatment failure. There is no restriction of CS usage after Day 210.

## 4.6.2 Other Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in APPENDIX 4. All medications taken within 30 days prior to screening must be recorded on the eCRF.


- 1. Prior exposure to BOS161721
- 2. Patients who have received treatment with anti-CD20 monoclonal antibodies within 24 weeks of screening
- 3. Patients who have received treatment with cyclophosphamide within the 24 weeks prior to screening
- 4. Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria within 4 weeks for oral use or 8 weeks for topical use of screening
- 5. Patients who are currently receiving or are scheduled to receive plasmapheresis or lymphapheresis therapy, or have received such therapy within 24 weeks prior to screening
- 6. Patients who have received any live vaccines within 30 days of screening. Note: Furthermore, live vaccines should not be used during the course of the study and within the 2 months following last dose. Other inactivated vaccines such as tetanus, etc., may be used according to local guidelines during treatment period
- 7. Patients who are scheduled or anticipated to have elective surgery during the course of the study
- 8. Initiation of new immunosuppressant or anti-malarial agent is not permitted. Note: Dose reduction or replacement may be allowed due to intolerability or shortage for patients on a stable dose prior to study initiation

## 4.7 Women of Childbearing Potential

WOCBP is defined as any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) and is not postmenopausal.

See Section 4.7.2 for detailed information regarding contraceptive requirements for WOCBP.

# **4.7.1 Determination of Menopause**

Menopause is defined as at least 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes. Women under the age of 55 years must have a documented serum FSH level > 40 mIU/mL at screening to confirm menopause.

### 4.7.2 Contraception

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks, due to the mean terminal ½ life of the study drug.

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks, due to the mean terminal ½ life of the study drug.

Investigators shall counsel WOCBP and men who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy.


Investigators shall advise WOCBP and men who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

Patients must agree to either complete abstinence, defined as a complete avoidance of heterosexual activity, or the use of 2 methods of highly effective contraception from the following:

- Male condoms with spermicide
- Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as 1 of the acceptable methods of contraception since they will not be receiving study drug.
- IUDs, such as ParaGard®
- Vasectomy

Note: Women who are abstinent while participating in the study must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the patient chooses to forego complete abstinence.

Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing.

#### 4.8 Deviation from Inclusion/Exclusion Criteria

Deviation from the inclusion or exclusion criteria will not be allowed. If deviation of inclusion/exclusion criteria is discovered after randomization, the investigator should contact the medical monitor for discussion. A decision will be made whether to allow a patient to continue or withdrawal from the study medication.

See Section 6.8 for additional details.

## 4.8.1 Patient Withdrawal and Replacement

See Section 5.5 for reasons for removal from the trial. Withdrawn patients may be replaced during the MAD part of the study after discussion between the principal investigator or designee and sponsor.

### 5 STUDY PROCEDURES

Refer to the eCRF completion guidelines for data collection requirements and documentation of study assessments/procedures.

## 5.1 Screening

Screening will be the same for both the MAD and POC portions of the study.


Screening will take place from Day -28 to Day -1, and assessments may be performed over more than 1 visit. Confirmation that the most current IRB/IEC approved informed consent form (ICF) has been signed must occur before any study-specific screening procedures are performed. Procedures that are part of standard of care are not considered study-specific procedures and may be performed prior to informed consent and used to determine eligibility.

All screened patients will be assigned a unique screening number. The screening number will include a 3-digit site number and a 4-digit sequential number to identify patients from the time of screening. Only eligible patients who are confirmed by central review as meeting the inclusion/exclusion criteria, listed in Section 4.4 and Section 4.5 respectively, will be enrolled in the study. Screened patients who drop out of the clinical study before randomization will be recorded as screen failures. If rescreening occurs, the site will assign a new screening number.

Specific procedures at the screening visit will include:

- Medical history documentation
- Review of inclusion and exclusion criteria
  - o Patient medical records must contain documentation of SLE diagnosis
  - o C-SSRS
- Concomitant medication documentation
- Demographics
- Full physical examination
- Vital signs
- Chest x-ray (a prior x-ray can be used if taken within 12 weeks of screening date)
- Laboratory evaluations (non-fasting):
  - o Hematology and clinical chemistry
  - o Serology (Hepatitis B and C; HIV-1/2 combination)
  - o TB test
  - o CRP
  - o Direct Coomb's test (if indicated for hemolytic anemia)
  - CD4+ count, total IgG and IgM levels, plasma
     CCI
  - Serum pregnancy test (WOCBP)
  - o FSH (postmenopausal women under age 55 years)
  - o Spot urine for protein/creatinine ratio
  - Urinalysis
  - Stool sample
- 12-lead ECG
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, Physician's Global Assessment (PGA) of disease activity

Screening procedures are listed in the Schedule of Assessments (Table 1 and Table 4), and details are provided in Section 6.


# 5.1.1 Retesting During Screening Period

A single retesting of laboratory parameters and/or other assessments during the screening period is permitted (in addition to any parameters that require a confirmatory value) only if:

- medically indicated
- there is evidence a laboratory sample was mislabeled, indeterminate, inadequately processed, and/or deteriorated in transit to the central laboratory

Any new result will override the previous result (ie, the most current result prior to randomization) and is the value by which study inclusion/exclusion will be assessed, as it represents the patient's most current clinical state. This will also apply to patients who are being rescreened.

# 5.2 Enrollment/Randomization and Day 0 Treatment

Randomization should occur after patient eligibility for enrollment has been confirmed by the central eligibility review. The central eligibility review team has the final decision on patient eligibility and can decide the patient is not eligible for the study based on their review of the eligibility packet.

Prior to randomization, the study site should confirm that the patient still meets inclusion/exclusion criteria (especially SLE disease activity and treatment). The site will obtain a randomization number when registering the patient in IWRS. All patients will receive BOS161721 or placebo according to the kit number assigned by the IWRS randomization scheme.

After randomization, procedures include:

- PROs: CCI
- C-SSRS
- Laboratory evaluations (fasting):
  - o Hematology and clinical chemistry
  - o Direct Coomb's test (if indicated for hemolytic anemia)
  - CD4+ count, total IgG and IgM levels, plasma CC , plasma CC and , whole blood for leukocyte immunophenotype (leukocyte immunophenotype for MAD patients only)
  - o ADA
  - o pSTAT3 (predose [trough] samples only in Phase 1b)
  - o CCI
  - o CCI
  - See Table 4 and Table 1 for details of PK sampling in the MAD and POC portions
  - o Urine pregnancy test will be collected on WOCBP prior to study drug administration


- o Spot urine for protein/creatinine ratio
- o Urinalysis
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Full physical examination
- Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours postdose on Day 0)
- 12-lead ECG (prior to PK blood draw)
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, PGA)
- SLICC/ACR damage index
- Study drug administration:
  - Administration of BOS161721 or placebo will take place on-site, and is discussed in Section 7.3
- Injection site reaction assessment performed at 2 hours postdose

Procedures on Day 0 are listed in the Schedule of Assessments (Table 1 and Table 4), and details are provided in Section 6.

All patients who are enrolled, randomized, and receive study drug, or undergo study-specific procedures should reconsent with any updated versions of IRB/IEC approved informed consents during study participation as applicable and per institutional guidelines.

## 5.3 Treatment Period/Follow-Up Visits

The following procedures will be performed as indicated in the Schedule of Assessments (Table 1 and Table 4). See Schedule of Assessment tables for allowable windows for each visit.

- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- PROs: CC
- Urine pregnancy tests will be collected on WOCBP prior to study drug administration
- Injection site reaction assessments will be performed predose
- Direct Coomb's test (if indicated for hemolytic anemia)
- Spot urine for protein to creatinine ratio
- Urinalysis
- · CCI
- Plasma CCI
- PGA, BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, and the CLASI will be completed
- SLICC/ACR Damage Index will be completed at Day 180
- C-SSRS


- ECGs prior to PK blood draw
- See Table 4 and Table 1 for details of PK sampling in the MAD and POC studies, respectively
- Fasting hematology and chemistry assessments
- The CD4+ count and total IgG and IgM levels
- Plasma CC and CC ADA, and whole blood for leukocyte immunophenotype (leukocyte immunophenotype for MAD patients only)
- pSTAT3 (predose [trough] samples only Phase 1b)
- nAb will be analyzed by central lab if patient is positive for ADA
- CRP
- CCI

## 5.4 Safety Follow-Up Visits

Safety follow-up visits will take place at Days 210, 240, and 270. These visits will include the following assessments as indicated in the Schedule of Assessments (Table 1 and Table 4):

- PROs: CC
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Injection site reactions
- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Spot urine for protein/creatinine ratio and urinalysis
- Concomitant medication documentation
- BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, and PGA
- Fasting clinical laboratory assessments (hematology and clinical chemistry)
- Direct Coomb's test (if indicated for hemolytic anemia)
- Plasma CCI
- CCI
- 12-lead ECG (prior to PK blood draw)
- CRP
- ADA
- CCI
- Urine pregnancy test
- See Table 4 and Table 1 for details of PK sampling in the MAD and POC portions, respectively

#### 5.5 Premature Discontinuation

While patients are encouraged to complete all study evaluations, they may withdraw from the study at any time and for any reason. Every effort will be made to determine why any patient


withdraws from the study prematurely. If the patient is unreachable by telephone, a registered letter, at the minimum, should be sent to the patient requesting him/her to contact the clinic.

All patients who withdraw from the study with an ongoing AE or SAE must be followed until the end of study or until the event is resolved or deemed stable, respectively.

If a patient withdraws prematurely after dosing, an end of treatment (EOT) visit should be performed (Day 180) and a last follow-up visit 90 days after dosing should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 5.4).

Patient participation may be terminated prior to completing the study and the reason recorded as follows:

- AE/SAE
- Protocol deviation
- Lost to follow-up
- Patient withdraws consent at their own request
- Investigator decision
- Decision by sponsor (other than AE/SAE, protocol deviation, or lost to follow-up)

Withdrawn patients may be replaced after discussion between the investigator or designee and sponsor.

#### 6 ASSESSMENTS

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances, outside of the control of the investigator, which may make it unfeasible to perform the test. In these cases, the investigator will take all steps necessary to ensure the safety and wellbeing of the patient. When a protocol required test cannot be performed the investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. All protocol violations are entered directly into the eCRFs.

# 6.1 Medical History, Demographic and Other Baseline Information

The medical history comprises:

- General medical history
- Documentation of SLE diagnosis
- Historical medication therapy for SLE

The following demographic information will be recorded:

Age


- Ethnic origin (Hispanic/Latino or not Hispanic/not Latino)
- Race (White, American Indian/Alaska Native, Asian, Native Hawaiian or other Pacific Islander, Black/African American)
- Height (without shoes, in cm)
- Body weight, without shoes (kg)
- BMI  $[kg/m^2]$

Other baseline characteristics will be recorded as follows:

- Concomitant medication documentation (see Section 4.6)
- Status of child bearing potential and contraception

# **6.2** Safety Assessments

### **6.2.1** Laboratory Assessments

Laboratory tests will be performed at times defined in the Schedule of Assessments (Table 1 and Table 4). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

A central laboratory will be used (with the exception of urine pregnancy tests) to ensure accuracy and consistency in test results. Laboratory/analyte results that could unblind the study (ie, biomarker results) will not be reported to investigative sites. Urinalysis will be performed on midstream, clean catch specimens. Some biomarkers listed above will not be drawn at some sites due to geographical logistical challenges. See the laboratory manual for details.

Endpoint analyses will be based on changes from baseline assessments at Days 120 and 210.

Table 2. Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| Hemoglobin | BUN | pН | Spot urine for protein/creatinine ratio |
| Hematocrit | Creatinine | Glucose (qual) | FSH <sup>b</sup> |
| RBC count | Glucose (fasting) | Protein (qual) | Urine pregnancy test <sup>c</sup> |
| RDW | Calcium | Blood (qual) | QuantiFERON®-TB Gold In-Tube test |
| MCV | Sodium | Ketones | (QFT-G) <sup>d</sup> |
| MCH | Potassium | Nitrites | Serology <sup>d</sup> (Hepatitis B and C; HIV-1/2 |
| MCHC | Chloride | Leukocyte esterase | combination) |
| Platelet count | Total CO <sub>2</sub> (bicarbonate) | Urobilinogen | Stool sample <sup>e</sup> |
| WBC count | AST, ALT | Urine bilirubin | Serum pregnancy test |
| CD4+ count | Total bilirubin | Microscopy <sup>a</sup> | |
| Total neutrophils | Alkaline phosphatase | | |
| (Abs) | Creatine kinase | | |
| Eosinophils (Abs) | Uric acid | | |
| Monocytes (Abs) | Albumin | | |
| Basophils (Abs) | Total cholesterol | | |
| Lymphocytes (Abs) | (fasting) | | |


**Table 2.** Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| | LDL-C (fasting) | | |
| | HDL-C (fasting) | | |
| | Triglycerides (fasting) | | |
| | Total protein | | |
| | PT/INR | | |
| | Additional Tests <sup>f</sup> | | Immunogenicity, PD and other |
| | (potential Hy's Law) | | <b>Biomarker Tests</b> |
| | AST, ALT (repeat) | | ADA |
| | Total bilirubin (repeat) | | $nAb^g$ |
| | Albumin (repeat) | | pSTAT3 (predose [trough] samples |
| | Alkaline phosphatase | | only in Phase 1b) |
| | (repeat) | | Total IgG & IgM |
| | Direct bilirubin | | Plasma CCI |
| | Indirect bilirubin | | Plasma CCI & CCI |
| | GGT | | Whole blood for leukocyte |
| | Prothrombin | | immunophenotype (for MAD patients |
| | time/international | | only) |
| | normalized ratio (repeat) | | CCI |
| | Creatine kinase (repeat) | | CCI |
| | | | CCI |
| | | | CRP |
| | | | Direct Coomb's test <sup>h</sup> |

Abbreviations: Abs = absolute; ADA = anti-drug antibody; ALT = alanine aminotransferase;

CC | ; CC | ; AST = aspartate aminotransferase; BUN = blood urea nitrogen; C = complement; CD4+ = cluster of differentiation 4; CRP = C-reactive protein;

CC | ;; FSH = follicle stimulating hormone;

GGT = gamma-glutamyltransferase; HDL-C = high-density lipoprotein cholesterol; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; INR = international normalized ration; IL-21 = interleukin 21; LDL-C = low-density lipoprotein cholesterol; MAD = multiple ascending doses;

ration; IL-21 = interleukin 21; LDL-C = low-density lipoprotein cholesterol; MAD = multiple ascending doses; MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = Mean corpuscular volume; nAb = neutralizing antibody; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; PT = prothrombin time; qual = qualitative; RBC = red blood cell; RDW = RBC distribution width; SAE = serious adverse event; SC = subcutaneous; CCl ; TB = tuberculosis.

- a. On all urine samples.
- b. At screening only, in women who are amenorrheic for at least 12 consecutive months and under 55 years old.
- c. For WOCBP.
- d. Screening only.
- <sup>e.</sup> At screening, and if a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- f. Additional testing for potential Hy's Law cases only (See Section 6.2.2.6.3).
- g. If patient is positive for ADA.
- h. If clinically indicated for hemolytic anemia.

### 6.2.1.1 Pregnancy testing

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or


continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, at the last follow up visit day (Day 270) and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures (see Section 5.4) are specified in the Schedule of Assessments (see Table 1 and Table 4).

See Section 6.2.2.7.1 for information on reporting of pregnancies as AEs/SAEs during the study.

### **6.2.1.2** Tuberculosis Screening

During the screening period, it must be determined and documented that a patient does not have evidence of active or latent or inadequately treated TB per the exclusion criteria (Section 4.5). The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).

### 6.2.1.2.1 Mycobacterium Tuberculosis Testing Using QuantiFERON Test<sup>40</sup>

QuantiFERON®-TB Gold In-Tube (QFT-G) is an *in vitro* diagnostic test using a peptide cocktail simulating ESAT-6, CFP-10, and TB 7.7 proteins to stimulate cells in heparinized whole blood. Detection of INFγ performed by enzyme-linked immunosorbent assay (ELISA) is used to identify *in vitro* responses to these peptide antigens that are associated with Mycobacterium tuberculosis infection. QFT-G is an indirect test for M. tuberculosis infection (including disease) and is intended for use in conjunction with risk assessment, radiography and other medical and diagnostic evaluations.

Test results will be reported as positive, negative, or indeterminate. A negative QFT-G test result is required to meet the inclusion criterion. In the case of an indeterminate result, repeat tests should be permitted for the purpose of determining eligibility of patients to enroll in this study. If a repeat test is indeterminate again, the patient is a screen failure. The procedure for using this test and interpreting the results will be described fully in the laboratory manual, which will be provided to investigators.

#### **6.2.2** Adverse Events

#### 6.2.2.1 Definitions

An AE is defined as any untoward medical occurrence experienced by a study patient, whether or not considered drug related by the principal investigator.

AEs are unfavorable changes in a general condition, subjective or objective signs or symptoms, worsening of pre-existing concomitant disease, and clinically significant abnormality in laboratory parameters observed in a patient in the course of a clinical study.


Non-serious SLE manifestations or abnormal laboratory results related to SLE disease activity would not be recorded as AEs unless they meet the definition for SAEs (Section 6.2.2.5).

# **6.2.2.2** Recording of Adverse Events

AEs should be collected and recorded for each patient from the date of the first dose of study drug until the end of their participation in the study, including the safety follow up period.

AEs may be volunteered spontaneously by the study patient, or discovered by the study staff during physical examinations or by asking an open, nonleading question such as 'How have you been feeling since you were last asked?' All AEs and any required remedial action will be recorded on the Adverse Events eCRF and Safety Adverse Event Form. The details of the AE, date of AE onset, date of AE outcome, and action taken for the AE will be documented together with the principal investigator's assessment of the seriousness of the AE and causal relationship to the study drug and/or the study procedure.

All AEs should be recorded individually, using diagnostic terms where possible. If the diagnosis is not established, individual symptoms may be reported. The AEs will subsequently be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

## **6.2.2.3** Severity of Adverse Events

Each AE will be assessed by the principal investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 criteria. <sup>41</sup> When changes in the severity (grade) of an AE occur more frequently than once a day, the maximum severity for the event should be noted for that day. Any change in severity of signs and symptoms over a number of days will be captured by recording a new AE, with the amended severity grade and the date (and time, if known) of the change.

### **6.2.2.4** Causality of Adverse Events

The principal investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (Table 3) should be selected based on medical judgment, considering the definitions below and all contributing factors.


| Table 3. | Causality | <b>Definitions</b> |
|-----------|-----------|--------------------|
| i able 3. | Causanty | Denninoi |

| Related | A clinical event, including laboratory test abnormality, occurs in a plausible time relationship to treatment administration and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (dechallenge <sup>a</sup> ) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge <sup>b</sup> procedure if necessary. |
|---|---|
| Unrelated | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative dechallenge and rechallenge information. Typically explained by extraneous factors (eg, concomitant disease, environmental factors, or other drugs or chemicals). |

- Dechallenge: Upon discontinuation of a drug suspected of causing an AE, the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation (positive dechallenge), or the symptoms continue despite withdrawal of the drug (negative dechallenge). Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia).
- Rechallenge: Upon re-administration of a drug suspected of causing an AE in a specific patient in the past, the AE recurs upon exposure (positive rechallenge), or the AE does not recur (negative rechallenge).

An unexpected adverse drug event is any adverse drug event for which the specificity or severity is not consistent with the current IP.

#### 6.2.2.5 Seriousness of Adverse Events

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life threatening; this means that the patient was at risk of death at the time of the event; it does not mean that the event hypothetically might have caused death if it were more severe
- Requires hospitalization or prolongation in existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly or birth defect
- Is other important medical event (see below)

Important medical events that do not result in death, are not life threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such events are:

- Intensive treatment in an emergency room or at home for allergic bronchospasm
- Blood dyscrasias or convulsions that do not result in inpatient hospitalization
- Development of drug dependency or drug abuse


Hospitalization for elective surgery or routine clinical procedures that are not the result of AE (eg, elective surgery for a pre-existing condition that has not worsened) need not be considered SAEs. If anything untoward is reported during the procedure, that occurrence must be reported as an AE, either 'serious' or 'nonserious' according to the usual criteria.

Suspected unexpected serious adverse reactions (SUSARs) are AEs that are associated with the use of the drug and are serious and unexpected.

## 6.2.2.6 Adverse Events of Special Interest

AEs of special interest in this study include the following:

- 1. Anaphylaxis and serious allergic reactions
- 2. Grades 2 to 5 injection site reaction, including erythema, pain, and induration (See APPENDIX 6)
- 3. Drug Induced Liver Injury (DILI) assessed following Hy's Law
- 4. Malignancy (not including basal cell carcinoma or squamous cell carcinoma of skin)
- 5. Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, disseminated herpes simplex, disseminated tuberculosis, *Aspergillus* sp., *Candida albicans*, *Coccidioides immitis*, *Cryptococcus neoformans*, *Cytomegalovirus*, *Histoplasma capsulatum*, *Isospora belli*, and *Polyomavirus JC polyomavirus*
- 6. Cryptosporidiasis

## 6.2.2.6.1 Anaphylaxis and Serious Allergic Reactions

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria.<sup>42</sup> In the event of anaphylactic reaction or severe/serious hypersensitivity/allergic reaction, the patient must discontinue IP and emergency resuscitation measures implemented. In case of other mild to moderate hypersensitivity reaction, depending on the severity, the investigator may manage in accordance with the standard-of-care.

Anaphylaxis is highly likely when any one of the following 3 criteria is fulfilled:

- 1. Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (eg, generalized hives, pruritus, or flushing, swollen lips-tongue-uvula) and at least 1 of the following:
  - a. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow [PEF], hypoxemia)
  - b. Reduced blood pressure or associated symptoms of end-organ dysfunction (eg, hypotonia [collapse], syncope, incontinence)
- 2. Two or more of the following that occur rapidly after exposure to a likely allergen for that patient (minutes to several hours):
  - a. Involvement of the skin-mucosal tissue (eg, generalized hives, itch-flush, swollen lips-tongue-uvula)


- b. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)
- c. Reduced blood pressure or associated symptoms (eg, hypotonia [collapse], syncope, incontinence)
- d. Persistent gastrointestinal symptoms (eg, crampy abdominal pain, vomiting)
- 3. Reduced blood pressure after exposure to known allergen for that patient (minutes to several hours):
  - a. Systolic blood pressure of less than 90 mm Hg or greater than 30% decrease from the patient's baseline

### **6.2.2.6.2 Injection Site Reactions**

Injection site reactions are to be captured and reported as AEs. These will include Grades 2 to 5 injection site erythema, pain, and induration (see APPENDIX 6), which are also captured as Adverse Events of Special Interest (See Section 6.2.2.6). The investigator should provide a clear description of the observed or reported AE including location and severity. All concomitant treatments used to treat injection site reactions should be recorded and captured in the eCRF, together with the AE of injection site reactions.

### 6.2.2.6.3 Potential Drug-Induced Liver Injury

Abnormal values in AST and/or ALT levels concurrent with abnormal elevations in total bilirubin level that meet the criteria outlined below in the absence of other causes of liver injury are considered potential cases of DILI, and as potential Hy's Law cases, and should always be considered important medical events. If symptoms compatible with DILI precede knowledge of serum chemical test abnormalities, liver enzyme measurements should be made immediately, regardless of when the next visit or monitoring interval is scheduled. In some cases, symptoms may be an early sign of injury and although typically less sensitive than serum enzyme elevations, they may indicate a need for prompt serum testing. An increase in liver enzymes should be confirmed by a repeated test within 48 to 72 hours following the initial test, prior to reporting of a potential DILI event. Patients will continue to have weekly or biweekly liver enzyme measurements until resolution or levels return to baseline.

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 6.2.2.7.2 for reporting details).

Potential DILI is defined as:

1. ALT or AST elevation  $> 3 \times ULN$ 

AND

2. Total bilirubin > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)

**AND** 


3. No other immediately apparent possible causes of ALT or AST elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic

The patient should return to the investigational site and be evaluated as soon as possible, include laboratory tests, detailed history, and physical assessment. In addition to repeating measurements of AST and ALT, laboratory tests should include albumin, CK, total bilirubin, direct and indirect bilirubin, GGT, prothrombin time (PT)/International Normalized Ratio (INR), and alkaline phosphatase. A detailed history, including relevant information, such as review of ethanol, acetaminophen, recreational drug and supplement consumption, family history, occupational exposure, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and work exposure, should be collected. Further testing for acute hepatitis A, B, or C infection and liver imaging (eg, biliary tract) may be warranted. All cases confirmed on repeat testing as meeting the laboratory criteria defined above, with no other cause for liver function test (LFT) abnormalities identified at the time should be considered potential Hy's Law cases irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal LFTs. Such potential Hy's Law cases should be reported as SAEs.

Study drug discontinuation is considered if there is marked serum AST or ALT elevation or evidence of functional impairment (as indicated by rising bilirubin or INR, which represent substantial liver injury) that is related to study drug. Discontinuation of treatment should be considered if:

- ALT or AST  $> 8 \times ULN$
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks

Discontinuation of treatment must occur if:

- ALT or AST >3 × ULN and (total bilirubin > 2 × ULN or INR > 1.5)
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%)

### 6.2.2.6.4 Malignancy

The identification of a malignancy event will be made by the study site and communicated to the sponsor or designee. AEs should be reported as serious per the criteria in Section 6.2.2.5.

After the first dose of study drug, when there is a decision to biopsy a potentially malignant tumor, lymph node, or other tissue (with the exception of suspected basal cell/squamous cell), the investigator and/or consultant(s) should contact the sponsor clinicians or designee to discuss the issue and any decisions as soon as possible. Basal cell carcinoma or squamous cell carcinoma of skin is not considered an AE of special interest.


#### 6.2.2.6.5 Specific Infections

Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, disseminated herpes simplex, disseminated tuberculosis, *Aspergillus* sp., *Candida albicans*, *Coccidioides immitis*, *Cryptococcus neoformans*, *Cytomegalovirus*, *Histoplasma capsulatum*, *Isospora belli*, or *Polyomavirus JC polyomavirus* will be recorded as AEs of special interest.

Cryptosporidiosis is also considered an AE of special interest. Patients will be evaluated for cryptosporidium in the stool at screening, and as clinically indicated (eg, watery diarrhea) during the study. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

## **6.2.2.7** Reporting of Adverse Events

AE reporting will be carried out in accordance with applicable local regulations, including regulatory agency and IRB reporting requirements.

Each AE is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

## **6.2.2.7.1** Reporting of Pregnancy

As information is available, a pregnancy diagnosed during the study will be reported within 24 hours to the sponsor via the Pregnancy Notification and Outcome Form, including pregnancy in female patients who received study drug and female partners of male study patients who received study drug. The pregnancy should be followed to term and/or outcome and this outcome should also be reported to the sponsor via the Pregnancy Notification and Outcome Form. Pregnancy itself is not regarded as an AE or SAE unless there is complication.

In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an AE or SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live born, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as serious


adverse events when the investigator assesses the neonatal death as related or possibly related to exposure to investigational product.

## **6.2.2.7.2** Reporting of Serious Adverse Events

The principal investigator is responsible for providing notification to the sponsor of any SAE via the Safety Adverse Event Form, whether deemed study drug related or not, that a patient experiences during their participation in this study within 24 hours of becoming aware of the event.

If an SAE is fatal or life threatening, notification to the sponsor must be made aware immediately, irrespective of the extent of available AE information. This timeframe also applies to additional new information (follow-up) on previously forwarded SAE reports as well as to the initial and follow-up reporting of exposure during pregnancy and exposure via breastfeeding cases. In the rare event that the investigator does not become aware of the occurrence of an SAE immediately (eg, if an outpatient study patient initially seeks treatment elsewhere), the investigator is to report the event within 24 hours after learning of it and document the time of his/her first awareness of the AE.

The principal investigator will review each SAE and evaluate the intensity and the causal relationship of the event to the study drug. All SAEs will be recorded from the time of first dose of study drug through the safety follow-up period (up to Day 270). SAEs occurring after the final follow-up visit and coming to the attention of the principal investigator must be reported only if there is (in the opinion of the principal investigator) reasonable causal relationship with the study drug.

As a minimum requirement, the initial notification should provide the following information:

- Study number
- Patient number
- Details of the SAE (verbatim details are sufficient for immediate notification)
- Criterion for classification as 'serious'
- Causality assessment (which may be updated in a follow-up report when sufficient information is available to make this classification)

Initial reports of SAEs must be followed later with detailed descriptions, including clear photocopies of other documents as necessary (eg, hospital reports, consultant reports, autopsy reports, etc), with the study patient's personal identifiers removed. All relevant information obtained by the principal investigator through review of these documents will be recorded and submitted to the sponsor within 24 hours of receipt of the information. If a new Safety Adverse Event Form is submitted, then the principal investigator must sign and date the form. The sponsor may also request additional information on the SAE, or clarification of omitted or discrepant information from the initial notification, which the principal investigator or an authorized delegate should submit to the sponsor within 24 hours of the request as possible.


# **6.2.2.7.3** Reporting of Adverse Events of Special Interest

AEs of special interest will be reported to safety immediately or within 24 hours of the site becoming aware of the event and recorded as such on the Adverse Events eCRF and Safety Adverse Event Form.

Potential DILI will be reported based on specifications mentioned in Section 6.2.2.6.3.

Each AE of special interest is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

## **6.2.2.8** Follow Up of Adverse Events

All AEs will be followed up through the safety follow-up visits. All SAEs experienced by a patient, irrespective of the suspected causality, will be monitored until the event has resolved, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the principal investigator and medical monitor, until there is a satisfactory explanation for the changes observed, or until the patient is lost to follow-up.

See Section 6.2.2.7.1 for details related to follow-up of pregnancy. See Section 6.2.2.6.3 for details related to follow-up of potential DILI. See Section 6.2.2.6.4 for details related to follow-up of malignancy.

# 6.2.3 Vital Signs

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (Table 1 and Table 4). Vital signs will be assessed on Day 0 at predose and at Day 0, 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq 5$  minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

## 6.2.4 12-Lead Electrocardiograms

ECG will be assessed as specified in the Schedule of Assessments (Table 1 and Table 4). ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

The ECG will include all 12 standard leads and a Lead II rhythm strip on the bottom of the tracing. The ECG will be recorded at a paper speed of 25 mm/second. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QT interval corrected for heart rate using Fridericia's formula (QTcF).


All ECGs must be evaluated by a qualified physician or qualified designee for the presence of abnormalities and will be captured electronically and retained for future evaluation if required, up to the time of the clinical study report (CSR) completion.

### 6.2.5 Physical Examinations

The full physical examination will be completed at screening and Day 0. It includes an assessment of general appearance and evaluation of head, eyes, ears, nose, mouth, throat, neck, thyroid, lymph nodes, and extremities, and dermatologic, respiratory, cardiovascular, gastrointestinal, musculoskeletal, neurologic, and psychiatric systems.

The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Table 1 and Table 4). It includes evaluation of patient complaints and SLE disease-related issues, and will exclude the genitourinary system.

## **6.2.6 C-SSRS**

The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed by Columbia University researchers for the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening.<sup>43</sup>

The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Table 1 and Table 4). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

#### **6.2.7** Injection Site Reactions

Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (Table 1 and Table 4). Local injection site reactions will be assessed at 2 hours postdose at baseline, and predose for each injection after baseline. Injection site reactions should be managed according to the standard of care. Injection site reactions, Grades 2 to 5, are to be reported as AEs of special interest (see Section 6.2.2.7.3).

#### 6.2.8 Immunogenicity

The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (Table 1 and Table 4). Blood samples (4 mL) to provide approximately 1.5 mL of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K<sub>2</sub>EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be


collected from all patients but only analyzed by a central lab if the patient had a positive ADA on Day 90.

After the first dose, if a patient tests positive in the validated confirmatory ADA assay, a sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay by a central lab.

## **6.3** Efficacy Assessments

All efficacy assessments will be performed at times defined in the Schedule of Assessments (Table 1 and Table 4).

#### **6.3.1 SLEDAI-2K**

The SLEDAI-2K is a validated instrument that measures disease activity in SLE patients at the time of the visit and in the previous 30 days. It is a global index and includes 24 clinical and laboratory variables that are weighted by the type of manifestation, but not by severity. The total score falls between 0 and 105, with higher scores representing increased disease activity. The SLEDAI-2K has been shown to be a valid and reliable disease activity measure in multiple patient groups. A SLEDAI -2K of 6 or more generally represents moderately to severely active disease. 44

#### 6.3.2 BILAG 2004

The BILAG-2004 index is an organ-specific 97-question assessment based on the principle of the doctor's intent to treat. Only clinical features attributable to SLE disease activity are to be recorded and based on the patient's condition in the last 4 weeks compared with the previous 4 weeks. It will be scored as not present (0), improved (1), the same (2), worse (3), or new (4). Disease activity is graded separately for 9 body systems to 5 different grades (A to E) as follows: A ("Active") is very active disease, B ("Beware") is moderate activity, C ("Contentment") is mild stable disease, D ("Discount") is inactive now but previously active, and E ("Excluded") indicates the organ was never involved. A shift from BILAG-2004 Grade A or B to a lower grade indicates a clinically relevant change in disease activity as the BILAG-2004 grades mirror the decision points for treatment interventions.

Only investigators that complete BILAG-2004 training will be allowed to perform the BILAG-2004 assessments. Preferably, the same investigator should evaluate the patient at each BILAG-2004 assessment from screening to study completion. The investigator must maintain documentation with descriptive details supporting the BILAG-2004 scoring (eg, chart, worksheet, clinic notes, and labs) at each visit.

See APPENDIX 5 for detailed specifications.

### 6.3.3 PGA of Disease Activity

The PGA is used to assess investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic


and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients". PGA worsening is defined as an increase of  $\geq$  30 mm from baseline.

When scoring the PGA, the assessor should always look back at the score from the previous visit.

### 6.3.4 Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response

### **6.3.4.1 SRI-4 Response**

The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. Response based on the SRI-4 is defined by:

1)  $\geq$  4-point reduction in SLEDAI-2K global score, 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B), and 3) no deterioration from baseline in the PGA by  $\geq$  30 mm. The SRI-4 response in patients with moderate to severe SLE is associated with broad improvements in clinical and patient-reported outcomes.<sup>45</sup>

## 6.3.4.2 SRI-5 and SRI-6 Response

Like the SRI-4, the SRI-5 and SRI-6 are composite indices of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. However, the SRI-5 and SRI-6 are computed with a minimal five-point or six-point improvement in SLEDAI-2K being required, respectively.<sup>46</sup>

### 6.3.4.3 BICLA Response

The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and PGA. BICLA response is defined as 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (eg, all B [moderate disease] scores falling to C [mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4)  $\leq$  10% deterioration in PGA score and 5) no treatment failure. 44 It is driven primarily by the BILAG, and has been used in Phase 2 and 3 mAb studies. 47

For the endpoints of BICLA response at Days 210, 240, and 270, patient scores will be completed and response determined.

### 6.3.5 CLASI Response

The CLASI is a comprehensive tool for assessment of disease activity and damage in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity. <sup>48</sup> Response is defined as 50% improvement from baseline in "A" or "B" scores. This assessment will be applied to all patients as all are required to have cutaneous disease activity.

For the secondary efficacy endpoint of CLASI response at Day 210, patient scores on MAD and POC studies will be compared with baseline for 50% improvement.


#### 6.3.6 ACR-28 Joint Count

The ACR-28 joint count will evaluate the number of tender and swollen joints in the shoulder, elbow, wrist, hand, knee joints. Joints of the feet are excluded.

#### 6.4 Other Variables

# 6.4.1 SLICC/ACR Damage Index

The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in patients with SLE regardless of cause, with demonstrated content, face, criterion, and discriminant validity. It will be performed on Days 0 and 180.

### 6.4.2 **PROs**

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the CCI and the CCI and will be assessed as specified in the Schedule of Assessments (Table 1 and Table 4).



#### 6.5 Pharmacokinetic Assessments

During the MAD Phase 1b (all sites) and POC Phase 2 (select sites only) parts of the study, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to Table 4 and Table 1.

Plasma concentrations of BOS161721 will be measured using a validated immunoassay. The PK parameters will be calculated from the plasma concentration actual time profiles.

# 6.6 Pharmacodynamic Assessments

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (Table 1 and Table 4) for each of the following parameters:

- pSTAT3 (predose [trough] samples only Phase 1b)
- Antibodies: CCl
- Plasma complement (CCI)


- Plasma CCI and CCI
- Whole blood for leukocyte immunophenotype (for MAD patients only)

## 6.7 Pharmacokinetic/Pharmacodynamic Relationship

Evidence of any PK/PD relationships will be evaluated between BOS161721 plasma concentrations and the available PD endpoints and biomarkers.

### **6.8** Protocol Deviations

Protocol deviations will be documented during the study.

## 7 STUDY DRUG MANAGEMENT

## 7.1 Description

#### 7.1.1 Formulation



Additional information regarding dose preparation will be provided in a separate Pharmacy Manual.

### 7.1.2 Storage

All supplies of BOS161721 or placebo must be stored in accordance with the manufacturer's instructions. BOS161721 or placebo will be stored in a securely locked area, accessible to authorized persons only, until needed for dosing.

Information regarding storage and dose preparation will be provided in a separate Pharmacy Manual.

# 7.2 Packaging and Shipment

Investigational medicinal products will be supplied by Boston Pharmaceuticals, Inc. Investigational medicinal products will be packaged and labeled according to applicable local and regulatory requirements.

#### 7.3 Dose and Administration

Details of dosing are provided in Section 3.1.


Each unit dose will be prepared by a qualified staff member. The vials of investigational product (IP) will appear identical and will have a "blinded" label on the vials that will state mg or placebo. When the site goes into the IWRS to request the patient kit(s), the IWRS will assign the appropriate number of kits (regardless of assignment to placebo or active treatment) per the dose (ie, CC). If a patient is randomized to the placebo arm, they will receive the matching number of kits.

The designated staff member (or designee under the direction of the designated staff member) will dispense BOS161721 or placebo for each patient according to the protocol, randomization list, and Pharmacy Manual, if applicable.

After receiving sponsor approval in writing, the investigational site is responsible for returning all unused or partially used BOS161721 or placebo to the sponsor or designated third party or for preparing BOS161721 or placebo for destruction via incineration.

Further details are found in a separate Pharmacy Manual.

## 7.4 Accountability

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Used investigational product returned to the pharmacy may be maintained in an ambient condition. Unused product should follow the instructions in the Pharmacy Manual. The used product that is returned should be marked as 'returned' and kept separate from the products not yet dispensed.

All dispensing and accountability records will be available for sponsor review after database lock procedures are completed. During safety monitoring, the drug accountability log will be reconciled with the products stored in the pharmacy.

# 7.5 Prohibited Concomitant Therapy

Prohibited concomitant medications are discussed in Section 4.6 and APPENDIX 4 and will be listed as protocol violations if taken when not permitted.

# 7.6 Compliance

Dosing will be performed by trained, qualified personnel designated by the principal investigator. The date and time of dosing will be documented on each dosing day. Comments will be recorded if there are any deviations from the planned dosing procedures.

### **8 STATISTICS**

The following analyses are planned:

• An IA will be performed during the last cohort of the MAD portion to determine dose selection for the POC part of the study.


- An additional analysis may be performed for the MAD portion of the study when all MAD patients have completed the safety follow-up or withdrawn from the study, and prior to final analysis. Data from the POC part of the study will be excluded from this additional analysis.
- The final analysis will be performed when all patients have completed the POC safety follow-up or withdrawn from the study.
- Safety analyses will be performed for DMC reviews throughout the study to evaluate dose escalation decisions and accumulating safety data. The frequency and details of the content and format of the safety review meetings will be described in the SAP and/or DMC charter.

All statistical analyses will be performed using Statistical Analysis Software (SAS®) Version 9 or higher.

The following standards will be applied for the analysis unless otherwise specified. Data will be summarized descriptively by treatment and overall for each study portion. For the MAD part of the study, BOS161721 will be summarized overall and by each dose level, and placebo patients from each cohort will be combined. Select parameters may be summarized using patients from both study parts. Statistical testing will be performed on data from the Phase 2 portion only.

Continuous data will be summarized using number, mean, standard deviation (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, median, and maximum. Categorical data will be summarized by treatment group using frequency tables (number and percentage). Time to event data will be summarized using counts, medians, 25<sup>th</sup> and 75<sup>th</sup> percentiles, and standard error. All data will be listed for all patients.

Statistical inference will be based on a 2-tailed test with an overall 0.10 level of significance, unless stated otherwise.

The effects of noncompliance, background therapy use, treatment discontinuations, premature withdrawal from study and covariates will be assessed to determine the impact on the general applicability of results from this study. Exploratory analyses of the data will be conducted as deemed appropriate. Any deviations from the planned analyses will be described and justified in the final integrated CSR.

Protocol deviations and prohibited medications that define medication failures will be fully assigned and documented before database lock and unblinding.

Further details of the analysis, including the handling of missing data, transformations and other data handling procedures will be provided in the SAP.

# 8.1 Sample Size

Sample size in the Phase 1b part of the study is based on operational consideration.

The sample size in the Phase 2 portion is based on the primary endpoint, SRI-4 Response at Day 210. Approximately 156 additional patients will be randomized in a 2:1 ratio to BOS161721 versus placebo to achieve 132 evaluable patients in the FAS. This assumes


24 patients will drop prior to having received treatment and an evaluable post-baseline efficacy measure. Enrollment and randomization will be monitored in a blinded fashion and increased if needed to ensure at least 132 patients are randomized into the FAS.

A total of 132 patients randomized provides more than 80% power to detect a treatment difference of 25% in SRI-4 response rates at Day 210, based on a targeted 2-sided significance level of 10% and using a 2-sided Pearson's chi-squared test. This assumes of a response rate of 65% for BOS161721 and 40% for placebo, where missing data at Day 210 is carried forward from most recent non-missing result and patients are treated as a non-responder if a prohibited medication defined as a medication failure occurs.

#### **8.2** Statistical Methods

# 8.2.1 Analysis Populations

The primary efficacy analysis will be based on the FAS, defined as all patients who receive at least 1 dose of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. FAS analyses will be conducted on the basis of the randomized treatment.

A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be identified based on blinded data prior to study unblinding. PP analyses will be conducted on the basis of the randomized treatment.

Safety analyses will be based on the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. Safety analyses will be conducted on the basis of actual treatment received.

Pharmacokinetic analysis will be conducted on the PK analysis set, defined as the FAS with sufficient concentration data for the calculation of PK parameters.

#### 8.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized using all randomized patients.

## 8.2.3 Primary Efficacy Endpoint(s)

The proportion of patients who achieve a SRI-4 response at Day 210 will be assessed via Pearson's chi-squared analysis. The primary efficacy endpoint will be analyzed using the FAS and if needed repeated in the PP analysis set. Missing values will be addressed by employing a last observation carried forward (LOCF) analysis. Other imputation methods may be employed as a sensitivity analysis and will be described in the SAP. Additional analyses exploring impact of baseline factors such as baseline disease severity, race, and other characteristics may be performed.

Patients that received prohibited medications or unallowable CS usage as described in Section 4.6 will be considered "medication failures" and will be treated as statistical


non-responders at time points on or following the first date of prohibited medication or unallowable CS usage for the primary efficacy analysis. The determination of medication failures will be reviewed using blinded data and finalized prior to unblinding.

The superiority of BOS161721 relative to placebo will be evaluated. If the proportion of SRI-4 responders for the selected POC dose in BOS161721 arm is higher than that of the placebo arm, then BOS161721 will be considered superior to placebo if the 2-sided p-value is less than 0.10. Secondary and exploratory endpoints for this POC portion will be evaluated based on the same statistical hypothesis.

#### 8.2.4 Secondary Efficacy Endpoint(s)

Binary efficacy endpoints will be assessed via Pearson's chi-squared analysis. Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) and treatment will be compared using the F-test. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test. The secondary efficacy endpoints will be analyzed on the FAS and if needed repeated in the PP analysis set. Details including handling of missing data and "medication failures" will be available in the SAP.

#### 8.2.5 Analysis of Safety

# 8.2.5.1 Safety Analysis

Safety analyses will be performed on the SS. AE data will be coded to system organ class and preferred term using MedDRA. The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term, will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be coded using the WHO Drug dictionary. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters will be summarized at each individual visit.

#### 8.2.6 Pharmacokinetic and Pharmacodynamic Data

#### 8.2.6.1 Analysis of Pharmacokinetic Data

PK parameters will be calculated from concentration data collected during the MAD Phase 1b portion of the study using non-compartmental analysis and include the following:

•  $C_{max}$ ,  $T_{max}$ , AUC,  $t_{\frac{1}{2}}$ , CL,  $V_d$ 

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:


• A listing of all plasma BOS161721 concentrations by patient at actual times post dose;

• A descriptive summary of plasma BOS161721 concentrations. Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.

#### 8.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Exploratory analyses examining the relationship between PD parameters and PK concentration and PK parameters will be performed.

#### 8.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints.

## 8.3 Interim Analysis and Power

One IA is planned for this study and will be conducted at the time of the POC decision for dose selection.

Since there is no IA during the POC part of the study, there is no impact on the type 1 error.

#### 9 ETHICS AND RESPONSIBILITIES

#### 9.1 Good Clinical Practice

The procedures set out in this protocol are designed to ensure that the sponsor and the principal investigator abide by the principles of the International Council for Harmonisation (ICH) guidelines on GCP and the Declaration of Helsinki (Version 2013). The clinical study also will be carried out in the keeping with national and local legal requirements (in accordance with US IND regulations [21 CFR 56]).

#### 9.2 **DMC**

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for BOS161721. The recommendations made by the DMC (ie, dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will


forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.

The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) suggest dose for POC portion of the study as described in Section 3.1.1.3.

The DMC considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

The DMC will have access to unblinded treatment information during the clinical trial. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of BOS161721 treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.

# 9.3 Institutional Review Board/Independent Ethics Committee

Independent Ethics Committees/IRB must meet the guidelines set out by the U.S. Food and Drug Administration (FDA) and conform to local laws and customs where appropriate. Written IRB/IEC approval for the protocol and the signed ICF must be obtained and transmitted to Boston Pharmaceuticals or representative before the study can be initiated. The IRB/IEC must be informed of and approve all protocol amendments. The investigator will ensure that this study is conducted in full conformance with all applicable local and regional laws and regulations. The complete text of the World Medical Association Declaration of Helsinki is given in APPENDIX 2.

#### 9.4 Informed Consent

Before each patient undergoes any protocol required assessments or procedure, the written informed consent will be obtained according to the regulatory and legal requirements of the participating country. As part of this procedure, the principal investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study patient should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The principal investigator or designee will provide the sponsor with a copy of the IRB-approved ICF prior to the start of the study.


The informed consent document must be signed and dated; 1 copy will be handed to the patient and the principal investigator will retain a copy as part of the clinical study records. The principal investigator will not undertake any investigation specifically required for the clinical study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented.

If the informed consent document is revised, it must be reviewed and approved by the responsible IRB/IEC. Patients currently enrolled may need to sign this revision (based on IRB/IEC requirements) and all future patients enrolled in the clinical study will be required to sign this revised ICF.

# 9.5 Records Management

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes. The principal investigator or designee will cooperate with the sponsor's representative(s) for the periodic review of study documents to ensure the accuracy and completeness of the data capture system at each scheduled monitoring visit.

Electronic consistency checks and manual review will be used to identify any errors or inconsistencies in the data. This information will be provided to the respective study sites by means of electronic or manual queries.

The principal investigator or designee will prepare and maintain adequate and accurate study documents (medical records, ECGs, AE and concomitant medication reporting, raw data collection forms, etc.) designed to record all observations and other pertinent data for each patient receiving BOS161721 or placebo.

The principal investigator will allow sponsor representatives, contract designees, authorized regulatory authority inspectors, and the IRB to have direct access to all documents pertaining to the study.

Electronic case report forms are required and should be completed for each randomized patient. It is the principal investigator's responsibility to ensure the accuracy, completeness, legibility, and timeliness of the data reported on the patients' eCRF. Electronic case report forms should be completed in a timely fashion to support the study timelines. Source documentation supporting the eCRF data should indicate the patient's participation in the study and should document the dates and details of study procedures, AEs, and patient status. The principal investigator or designated representative should complete and the principal investigator should verify the source documents as the information is collected. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the Sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes.


#### 9.6 Source Documentation

The documents that will form the source data for the clinical study (eg, patient charts, laboratory reports) must be defined and documented in the in-house study master file prior to the start of the study. Data on the eCRFs which will be checked against source data during monitoring visits must also be defined and documented in the in-house study master file including the percentage of each of the source data to be verified and the percentage of patients' eCRFs to be monitored.

# 9.7 Study Files and Record Retention

According to ICH guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of BOS161721. However, these documents should be retained for a longer period if required by the applicable legal requirements.

#### 10 AUDITING AND MONITORING

Throughout the course of the study, the study monitor will make frequent contacts with the investigator. This will include telephone calls and on-site visits. The study will be routinely monitored to ensure compliance with the study protocol and the overall quality of data collected. During the on-site visits, the eCRFs will be reviewed for completeness and adherence to the protocol. As part of the data audit, source documents will be made available for review by the study monitor. The study monitor may periodically request review of the investigator study file to assure the completeness of documentation in all respects of clinical study conduct. The study monitor will verify that each patient has proper consent documentation from the patient and/or patient's authorized representative for study procedures and for the release of medical records to the sponsor, FDA, other regulatory authorities, and the IRB. The study monitor will also verify that assent was obtained for patients not capable of providing informed consent or that documentation is provided by the investigator explaining why the patient was unable to provide assent. The investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the investigator will permit inspection of the study files by authorized representatives of the regulatory agencies. On completion of the study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

Throughout the course of the study, the medical monitor will determine eligibility of all screened patients, will address any medical issues that might arise, clarify medical questions, review patient safety data (eg, AE/SAE, laboratory, and ECG), and partner with the study team in the overall study management. The study medical monitoring plan will document additional details of the study medical oversight and monitoring.

#### 11 AMENDMENTS

Protocol modifications, except those intended to reduce immediate risk to study patients, may be made only by Boston Pharmaceuticals. A protocol change intended to eliminate an apparent


immediate hazard to patients may be implemented immediately, provided the IRB/IEC is notified within 5 days.

Any permanent change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB/IEC and the investigator must await approval before implementing the changes. Boston Pharmaceuticals will submit protocol amendments to the appropriate regulatory authorities for approval.

If in the judgment of the IRB/IEC, the investigator, and/or Boston Pharmaceuticals, the amendment to the protocol substantially changes the study design and/or increases the potential risk to the patient and/or has an impact on the patient's involvement as a study participant, the currently approved written ICF will require similar modification. In such cases, informed consent will be renewed for patients enrolled in the study before continued participation.

#### 12 STUDY REPORT AND PUBLICATIONS

Boston Pharmaceuticals is responsible for preparing and providing the appropriate regulatory authorities with clinical study reports according to the applicable regulatory requirements.

By signing the protocol, the principal investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the principal investigator's name, address, qualifications, and extent of involvement.

The principal investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted and obtained approval from the sponsor in advance.

#### 13 STUDY DISCONTINUATION

Both Boston Pharmaceuticals and the principal investigator reserve the right to terminate the study at the investigator's site at any time. Should this be necessary, Boston Pharmaceuticals or a specified designee will inform the appropriate regulatory authorities of the termination of the study and the reasons for its termination, and the principal investigator will inform the IRB/IEC of the same. In terminating the study Boston Pharmaceuticals and the principal investigator will assure that adequate consideration is given to the protection of the patients' interests.

#### 14 CONFIDENTIALITY

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from Boston Pharmaceuticals, except to the extent necessary to obtain informed consent from patients who wish to participate in the trial or to comply with regulatory requirements. However, authorized regulatory officials, IRB/IEC personnel, Boston Pharmaceuticals, and its authorized representatives are allowed full access to the records.

Identification of patients and eCRFs shall be by initials, birthdate, or patient number. Documents that identify the patient (eg, the signed informed consent document) must be


maintained in confidence by the principal investigator. If required, the patient's full name may be made known to an authorized regulatory agency or other authorized official.


## 15 REFERENCES

1 Urowitz MB, Gladman DD. How to improve morbidity and mortality in systemic lupus erythematosus. Rheumatology 2000;39:238-44.

- 2 Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, et al. Morbidity and Mortality in Systemic Lupus Erythematosus During a 10-Year Period. Medicine 2003;82(5):299-308.
- 3 Pons-Estel GJ, Alarcón GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010;39(4):257. Epub 2009 Jan 10.
- 4 Kanta H, Mohan C. Three Checkpoints in lupus development: central tolerance in adaptive immunity, peripheral amplification by innate immunity, and end-organ inflammation. Genes and Immunity 2009;10:390-6.
- 5 Dall'Aqua WF, Kiener PA, Wu H. Properties of Human IgG1s Engineered for Enhanced Binding to the Neonatal Fc Receptor (FcRn). J Biol Chem. 2006 Aug 18, 281(33):23514-24.
- 6 Spolski R, Leonard WJ. The Yin and Yang of interleukin-21 in allergy, autoimmunity and cancer. Curr Opin Immunol. 2008a;20:295-301.
- 7 Asao H, Okuyama C, Kumaki S, Ishii N, Tsuchiya S, Foster D, et al. Cutting edge: the common gamma-chain is an indispensable subunit of the IL-21 receptor complex. J Immunol. 2001;167:1-5.
- 8 Habib T, Senadheera S, Weinberg K, Kaushansky K. The common gamma chain (gamma c) is a required signaling component of the IL-21 receptor and supports IL-21-induced cell proliferation via JAK3. Biochemistry. 2002;41:8725-31.
- 9 Spolski R, Leonard WJ. Interleukin-21: basic biology and implications for cancer and autoimmunity. Annu Rev Immunol. 2008b;26:57-79.
- 10 Puga I, Cols M, Barra CM, He B, Cassis L, Gentile M, et al. B-cell-helper neutrophils stimulate the diversification and production of immunoglobulin in the marginal zone of the spleen. Nat Immunol. 2011;13(2):170-80.
- 11 Costanzo A, Chimenti MS, Botti E, Caruso R, Sarra M, Monteleone G. IL-21 in the pathogenesis and treatment of skin diseases. J Dermatol Sci. 2010;60(2):61-6.
- 12 Avery DT, Bryant VL, Ma CS, de Waal Malefy R, Tangye SG. IL-21-induced isotype switching to IgG and IgA by human naive B cells is differentially regulated by IL-4. J Immunol. 2008;181:1767-79.
- 13 Rasmussen TK, Andersen T, Bak, RO, Yiu G, Sorensen CM, Stengaard-Pedersen K, et al. Overexpression of microRNA-155 increases IL-21 mediated STAT3 signaling and IL-21 production in systemic lupus erythematosus. Arthritis Research & Therapy 2015;17(154)


- 14 Ettinger R, Kuchen S, Lipsky PE. The role of IL-21 in regulating B-cell function in health and disease. Immunol Rev. 2008;223:60-86.
- 15 Caprioli F, Sarra M, Caruso R, Stolfi C, Fina D, Sica G, et al. Autocrine regulation of IL-21 production in human T lymphocytes. J Immunol. 2008;180(3):1800-7.
- 16 Yang L, Anderson DE, Baecher-Allan C, Hastings WD, Bettelli E, Oukka M, et al. IL-21 and TGF-beta are required for differentiation of human T(H)17 cells. Nature. 2008;454(7202):350-2.
- 17 Tangye SG, Ma CS, Brink R, Deenick EK. The good, the bad and the ugly TFH cells in human health and disease. Nat Rev Immunol. 2013;13(6):412-26.
- 18 Fantini MC, Rizzo A, Fina D, Caruso R, Becker C, Neurath MF, et al. IL-21 regulates experimental colitis by modulating the balance between Treg and Th17 cells. Eur J Immunol. 2007;37(11):3155-63.
- 19 Peluso I, Fantini MC, Fina D, Caruso R, Boirivant M, MacDonald TT, et al. IL-21 counteracts the regulatory T-cell-mediated suppression of human CD4+ T lymphocytes. J Immunol. 2007;178(2):732-9.
- 20 Hippen KL, Bucher C, Schirm DK, Bearl AM, Brender T, Mink KA, et al. Blocking IL-21 signaling ameliorates xenogeneic GVHD induced by human lymphocytes. Blood. 2012;119(2):619-28.
- 21 Davis ID, Skrumsager BK, Cebon J, Nicholaou T, Barlow JW, Moller NP, et al. An open-label, two-arm, phase I trial of recombinant human interleukin-21 in patients with metastatic melanoma. Clin Cancer Res. 2007;13:3630-6.
- 22 Frederiksen KS, Lundsgaard D, Freeman JA, Hughes SD, Holm TL, Skrumsager BK, et al. IL-21 induces in vivo immune activation of NK cells and CD8(+) T-cells in patients with metastatic melanoma and renal cell carcinoma. Cancer Immunol Immunother. 2008;57(10):1439-49.
- 23 Karrich JJ, Jachimowski LC, Nagasawa M, Kamp A, Balzarolo M, Wolkers MC, et al. IL-21- stimulated human plasmacytoid dendritic cells secrete granzyme B, which impairs their capacity to induce T-cell proliferation. Blood. 2013;121(16):3103-11.
- 24 Lindner S, Dahlke K, Sontheimer K, Hagn M, Kaltenmeier C, Barth TF, et al. Interleukin-21-induced granzyme B-expressing B-cells infiltrate tumors and regulate T-cells. Cancer Res. 2013;73(8):2468-79.
- 25 Monteleone G, Caruso R, Fina D, Peluso I, Gioia V, Stolfi C, et al. Control of matrix metalloproteinase production in human intestinal fibroblasts by interleukin 21. Gut. 2006;55(12):1774-80.
- 26 Nakou M, Papadimitraki ED, Fanouriakis A, Bertsias GK, Choulaki C, Goulidaki N, et al. Interleukin-21 is increased in active systemic lupus erythematosus patients and contributes to the generation of plasma B-cells. Clin Exp Rheumatol. 2013;31(2):172-9.


- 27 Li Q, Liu Z, Dang E, Jin L, He Z, Yang L, et al. Follicular helper T-cells (Tfh) and IL-21 involvement in the pathogenesis of bullous pemphigoid. PLoS One. 2013;8(7):e68145.
- 28 Liu R, Wu Q, Su D, Che N, Chen H, Geng L, et al. A regulatory effect of IL-21 on T follicular helper-like cell and B-cell in rheumatoid arthritis. Arthritis Res Ther. 2012;14(6):R255.
- 29 Kang KY, Kim HO, Kwok SK, Ju JH, Park KS, Sun DI, et al. Impact of interleukin-21 in the pathogenesis of primary Sjögren's syndrome: increased serum levels of interleukin-21 and its expression in the labial salivary glands. Arthritis Res Ther. 2011;13(5):R179.
- 30 Terrier B, Geri G, Chaara W, Allenbach Y, Rosenzwajg M, Costedoat-Chalumeau N, et al. Interleukin-21 modulates Th1 and Th17 responses in gianT-cell arteritis. Arthritis Rheum. 2012a;64(6):2001-11.
- 31 Terrier B, Costedoat-Chalumeau N, Garrido M, Geri G, Rosenzwajg M, Musset L, et al. Interleukin 21 correlates with T-cell and B-cell subset alterations in systemic lupus erythematosus. J Rheumatol. 2012b;39(9):1819-28.
- 32 International Conference on Harmonisation. Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals S6 (R1). 2011.
- 33 Wang W, Wang EQ, Balthasar JP. Monoclonal Antibody Pharmacokinetics and Pharmacodynamics. Clin Pharm & Ther 2008; 84(5):548-58.
- 34 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 35 Elsaesser H, Sauer K, Brooks DG. IL-21 is required to control chronic viral infection. Science. 2009;324(5934):1569-72
- 36 Kotlarz D, Zietara N, Uzel G, Weidemann T, Braun CJ, Diestelhorst J, et al. Loss-of-function mutations in the IL-21 receptor gene cause a primary immunodeficiency syndrome. J Exp Med. 2013;210(3):433-43.
- 37 Hunter PR, Nichols G. Epidemiology and clinical features of Cryptosporidium infection in immunocompromised patients. Clinical microbiology reviews. 2002;15(1):145-54.
- 38 Desjardins M, Mazer BD. B-cell memory and primary immune deficiencies: interleukin-21 related defects. Curr Opin Allergy Clin Immunol. 2013;13(6):639-45.
- 39 Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. *Nephron*. 1976;16(1):31-41.


- 40 Guidelines for Using the QuantiFERON®-TB Gold Test for Detecting Mycobacterium tuberculosis Infection, US: http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5415a4.htm.
- 41 NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, available at https://evs.nci.nih.gov/ftp1/CTCAE/About.html.
- 42 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 43 Posner K, Melvin G a, Stanley B, Oquendo M a, Gould M. Factors in the assessment of suicidality in youth. *CNS Spectr*. 2007;12(2):156-162.
- 44 Castrejon I, Tani C, Jolly M, Huang A, Mosca M. Indices to assess patients with systemic lupus erythematosus in clinical trials, long-term observational studies, and clinical care. Clin Exp Rheumatol 2014; 32(85):S85-95.
- 45 Furie R, Wang L, Drappa J, Illei G. Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] Response Is Associated with Global Benefit in Patients with Moderate to Severe SLE [abstract]. *Arthritis Rheumatol.* 2016; 68 (suppl 10).
- 46 Thanou A, Chakravarty E, James JA, Merrill JT. Which outcome measures in SLE clinical trials best reflect medical judgment? Lupus Science & Medicine 2014;1:e000005. doi:10.1136/lupus-2013-000005.
- 47 Wallace DJ, Kalunian K, Petri MA, Strand V, Houssiau FA, Pike M, et al. Efficacy and safety of epratuzumab in patients with moderate/severe active systemic lupus erythematosus: results from EMBLEM, a phase IIb, randomised, double-blind, placebo-controlled, multicentre study. *Ann Rheum Dis* 2014;73:183-90.
- 48 Albrecht J, Taylor L, Berlin JA, Dulay S, Ang G, Fakharzadeh S. The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index): An Outcome Instrument for Cutaneous Lupus Erythematosus. J Invest Derm. 2005;125(5):889-94.
- 49 Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is Valid, and Renal and Pulmonary Organ Scores are Predictors of Sever Outcome in Patients with Systemic Lupus Erythematosus. Br J Rheumatol. 1996;35:248-54.

50 **CC** 


# 16 APPENDICES

# APPENDIX 1 NAMES OF STUDY PERSONNEL




# APPENDIX 2 DECLARATION OF HELSINKI

# WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI

Ethical Principles
For
Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly
Helsinki, Finland, June 1964
and amended by the
29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
and the

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### A. INTRODUCTION

The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.

It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.

The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my subject will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the subject's interest when providing medical care which might have the effect of weakening the physical and mental condition of the subject."

Medical progress is based on research, which ultimately must rest in part on experimentation involving human subjects.

In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.

The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic, and therapeutic procedures and the understanding of the etiology and pathogenesis of disease. Even the best-proven prophylactic, diagnostic, and therapeutic methods must continuously be challenged through research for their effectiveness, efficiency, accessibility, and quality.

In current medical practice and in medical research, most prophylactic, diagnostic, and therapeutic procedures involve risks and burdens.


Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.

Research investigators should be aware of the ethical, legal, and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal, or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### B. BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.

Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.

Appropriate caution must be exercised in the conduct of research, which may affect the environment, and the welfare of animals used for research must be respected.

The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any SAEs. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.

The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles enunciated in this Declaration.

Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a subject of the research, even though the subject has given consent.

Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.


Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.

Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.

Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.

The subjects must be volunteers and informed participants in the research project.

The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the subject's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.

In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.

When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.

For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the investigator must obtain informed consent from the legally authorized representative in accordance with applicable law. These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.

When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the investigator must obtain that assent in addition to the consent of the legally authorized representative.

Research on individuals from whom it is not possible to obtain consent, including proxy or advance consent, should be done only if the physical/mental condition that prevents obtaining informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the


review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.

Both authors and publishers have ethical obligations. In publication of the results of research, the investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic, or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the subjects who are research subjects.

The benefits, risks, burdens, and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic, or therapeutic method exists.

At the conclusion of the study, every subject entered into the study should be assured of access to the best-proven prophylactic, diagnostic, and therapeutic methods identified by the study.

The physician should fully inform the subject which aspects of the care are related to the research. The refusal of a subject to participate in a study must never interfere with the subject-physician relationship.

In the treatment of a subject, where proven prophylactic, diagnostic, and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the subject, must be free to use unproven or new prophylactic, diagnostic, and therapeutic measures, if in the physician's judgment it offers hope of saving life, re-establishing health, or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases, new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.


# APPENDIX 3 COMMONLY USED CORTICOSTEROID EQUIVALENTS

| Medication | Prednisone Dose Equivalence |
|--------------------|-----------------------------|
| Prednisone | 1 mg |
| Cortisone | 5 mg |
| Hydrocortisone | 4 mg |
| Prednisolone | 1 mg |
| Methylprednisolone | 0.8 mg |
| Triamcinolone | 0.8 mg |
| Budesonide | 0.25 mg |
| Dexamethasone | 0.16 mg |
| Bethamethasone | 0.16 mg |


# APPENDIX 4 MEDICATION WASHOUT PERIODS

# WASHOUT TIMES OF MEDICATIONS BASED ON 5 HALF-LIVES

| Medication | <b>Discontinuing Prior to Signing Consent</b> |
|---|---|
| Abatacept (CTLA4Ig) | 24 weeks |
| Alefacept | 12 weeks |
| AMG 623 (blisibimod) | 24 weeks |
| Anifrolumab | 12 weeks |
| Atacicept (TACI-Ig) | 12 weeks |
| Belimumab | 24 weeks |
| Cyclophosphamide | 24 weeks |
| Cyclosporine (except for CSA eye drops) | 4 weeks for oral and 8 weeks for topical |
| Danazol | 4 weeks |
| Dapsone | 4 weeks |
| Eculizumab | 12 weeks |
| Efalizumab | 12 weeks |
| Epratuzumab | 24 weeks |
| Intravenous globulin | 4 weeks |
| Leflunomide | 8 weeks (4 weeks for washout with |
| | cholestyramine) |
| Lenalidomide with cholestiramine | 8 weeks |
| Lupuzor | 12 weeks |
| Memantine | 4 weeks |
| Natalizumab | 24 weeks |
| Ocrelizumab | 48 weeks (or 24 weeks with recovery of B cell) |
| Pimecrolimus | 4 weeks |
| Plasmapheresis | 24 weeks |
| Retinoids (oral or topical) | 4 weeks |
| Rituximab | 48 weeks (or 24 weeks with recovery of B cell) |
| Sirolimus | 4 weeks |
| Tacrolimus | 4 weeks |
| Thalidomide | 8 weeks |
| Tocilizumab | 12 weeks |


# APPENDIX 5 BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA)




# APPENDIX 6 INJECTION SITE REACTION GRADING SCALE

| Adverse event<br>Injection site reaction | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade<br>5 |
|---|---|---|---|---|---|
| Definition: A disorder<br>characterized by an<br>intense adverse reaction<br>(usually immunologic)<br>developing at the site of<br>an injection | Tenderness with<br>or without<br>associated<br>symptoms (eg,<br>warmth,<br>erythema,<br>itching) | Pain;<br>Lipodystrophy;<br>Edema;<br>phlebitis | Ulceration or<br>necrosis;<br>Severe tissue<br>damage;<br>Operative<br>intervention<br>indicated | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>indicated | Death |
| Pain | Mild pain | Moderate pain;<br>limiting<br>instrumental ADL | Severe pain;<br>limiting self-<br>care ADL | - | - |
| Rash<br>maculopapular/Erythema<br>/Induration | Macules/papules<br>covering <10%<br>BSA with or<br>without | Macules/papules<br>covering 10% -<br>30% BSA with or<br>without symptoms | Macules/papul<br>es covering<br>> 30% BSA<br>with or | - | - |
| Definition: A disorder<br>characterized by the<br>presence of macules<br>(flat) and papules<br>(elevated). Also known<br>as morbilliform rash, it is | symptoms (eg,<br>pruritus, burning,<br>tightness)<br>Erythema<br>covering <10%<br>BSA with or | (eg, pruritus,<br>burning, tightness);<br>limiting<br>instrumental ADL;<br>Erythema 30%<br>BSA with or | without<br>associated<br>symptoms;<br>limiting<br>self-care ADL | | |
| one of the most common<br>cutaneous adverse<br>events, frequently<br>affecting the upper trunk,<br>spreading centripetally,<br>and associated with | without<br>symptoms (eg,<br>pruritus, burning,<br>tightness) | without symptoms<br>(eg, pruritus,<br>burning, tightness);<br>limiting<br>instrumental ADL | Erythema covering > 30% BSA with or without associated | | |
| pruritus. | | | symptoms;<br>limiting<br>self-careADL | | |

ADL = active daily living


# APPENDIX 7 OPIOID ORAL MORPHINE MILLIGRAM EQUIVALENTS OF COMMONLY USED OPIOIDS

| Opioid | 30 mg morphine equivalent |
|----------------------|---------------------------|
| butorphanol | 4.3 mg/day |
| codeine | 200 mg/day |
| dihydrocodeine | 120 mg/day |
| fentanyl transdermal | 12.5 mg/day |
| hydrocodone | 30 mg/day |
| hydromorphone | 7.5 mg/day |
| levorphanol tartrate | 2.7 mg/day |
| meperidine HCl | 300 mg/day |
| oxycodone | 20 mg/day |
| oxymorphone | 10 mg/day |
| pentazocine | 81.1 mg/day |
| tapentadol | 75 mg/day |
| tramadol | 300 mg/day |

Note that this list is not comprehensive. If an opioid is being used which is not in this list, please see the appropriate conversion factor below.


## Opioid Oral Morphine Equivalent Conversion Factors<sup>a,b</sup>

| Type of Opioid (strength in units) | MME Conversion Factor |
|---|---|
| Buprenorphine film/table <sup>c</sup> (mg) | 30 |
| Buprenorphine patch <sup>d</sup> (mcg/hr) | 12.6 |
| Buprenorphine film (mcg) | 0.03 |
| Butorphanol (mg) | 7 |
| Codeine (mg) | 0.15 |
| Dihydrocodeine (mg) | 0.25 |
| Fentanyl buccal or SL tablets, or lozenge/troche <sup>e</sup> (mcg) | 0.13 |
| Fentanyl film or oral spray <sup>f</sup> (mcg) | 0.18 |
| Fentanyl nasal spray <sup>g</sup> (mcg) | 0.16 |
| Fentanyl patch <sup>h</sup> (mcg) | 7.2 |
| Hydrocodone (mg) | 1 |
| Hydromorphone (mg) | 4 |
| Levorphanol tartrate (mg) | 11 |
| Meperidine hydrochloride (mg) | 0.1 |
| Methadone <sup>i</sup> (mg) | 3 |
| > 0, \le 20 | 4 |
| > 20, ≤ 40 | 8 |
| > 40, ≤ 60 | 10 |
| > 60 | 12 |
| Morphine (mg) | 1 |
| Opium (mg) | 1 |
| Oxycodone (mg) | 1.5 |
| Oxymorphone (mg) | 3 |
| Pentazocine (mg) | 0.37 |
| Tapentadol <sup>j</sup> (mg) | 0.4 |
| Tramadol (mg) | 0.1 |

CDC = Centers for Disease Control; CMS = Centers for Medicare and Medicaid Services; FDA = Food and Drug Administration; MAT = Medication Assisted Treatment; MME = morphine milligram equivalent; OMS = Overutilization Monitoring System.

- a. The MME conversion factor is intended only for analytic purposes where prescription data is used to calculate daily MME. It is to be used in the formula: Strength per Unit × (Number of Units/Days Supply) × MME conversion factor = MME/Day. This value does not constitute clinical guidance or recommendations for converting patients from one form of opioid analgesic to another. Please consult the manufacturer's full prescribing information for such guidance. Use of this file for the purposes of any clinical decision-making warrants caution.
- b. National Center for Injury Prevention and Control. CDC compilation of benzodiazepines, muscle relaxants, stimulants, zolpidem, and opioid analgesics with oral morphine milligram equivalent conversion factors, 2016 version. Atlanta, GA: Centers for Disease Control and Prevention; 2016. Available at <a href="https://www.cdc.gov/drugoverdose/media/">https://www.cdc.gov/drugoverdose/media/</a>. For more information, send an email to Mbohm@cdc.gov.
- c. Buprenorphine formulations with a FDA approved indication for MAT are excluded from Medicare's Overutilization Monitoring System's opioid overutilization reporting.


- d. The MME conversion factor for buprenorphine patches is based on the assumption that 1 milligram of parenteral buprenorphine is equivalent to 75 milligrams of oral morphine and that one patch delivers the dispensed micrograms per hour over a 24 hour day. Example: 5 μg/hr buprenorphine patch × 24 hrs = 120 ug/day buprenorphine = 0.12 mg/day = 9 mg/day oral MME. In other words, the conversion factor not accounting for days of use would be 9/5 or 1.8.
  However, since the buprenorphine patch remains in place for 7 days, we have multiplied the conversion factor by 7 (1.8 × 7 = 12.6). In this example, MME/day for 4 5 μg/hr buprenorphine patches dispensed for use over 28 days would work out as follows: Example: 5 μg/hr buprenorphine patch × (4 patches/28 days) × 12.6 = 9 MME/day. Please note that because this allowance has been made based on the typical dosage of 1 buprenorphine patch per 7 days, you should first change all Days Supply in your prescription data to follow this standard, i.e., Days Supply for buprenorphine patches = number of patches x 7.
- e. The MME conversion factor for fentanyl buccal tablets, sublingual tablets, and lozenges/troche is 0.13. This conversion factor should be multiplied by the number of micrograms in a given tablet or lozenge/troche.
- f. The MME conversion factor for fentanyl film and oral spray is 0.18. This reflects a 40% greater bioavailability for films compared to lozenges/tablets and 38% greater bioavailability for oral sprays compared to lozenges/tablets.
- g. The MME conversion factor for fentanyl nasal spray is 0.16, which reflects a 20% greater bioavailability for sprays compared to lozenges/tablets.
- h. The MME conversion factor for fentanyl patches is based on the assumption that 1 milligram of parenteral fentanyl is equivalent to 100 milligrams of oral morphine and that 1 patch delivers the dispensed micrograms per hour over a 24 hour day. Example:  $25 \,\mu g/hr$  fentanyl patch  $\times$  24 hrs = 600 ug/day fentanyl = 60 mg/day oral morphine milligram equivalent. In other words, the conversion factor not accounting for days of use would be 60/25 or 2.4. However, since the fentanyl patch remains in place for 3 days, we have multiplied the conversion factor by  $3 \, (2.4 \times 3 = 7.2)$ . In this example, MME/day for  $10 \, 25 \, \mu g/hr$  fentanyl patches dispensed for use over 30 days would work out as follows:
  - Example:  $25 \mu g/hr$  fentanyl patch  $\times$  (10 patches/30 days)  $\times$  7.2 = 60 MME/day. Please note that because this allowance has been made based on the typical dosage of 1 fentanyl patch per 3 days, you should first change all Days Supply in your prescription data to follow this standard, i.e., Days Supply for fentanyl patches = number of patches  $\times$  3.
- i. The CDC MME conversion factor to calculate morphine milligram equivalents is 3. CMS uses this conversion factor when analyzing Medicare population opioid use. CMS uses the graduated methadone MME conversion factors to calculate MME within the OMS for identifying and reporting potential opioid overutilizers. https://www.cdc.gov/drugoverdose/pdf/calculating total daily dose-a.pdf.
- j. Tapentadol is a mu receptor agonist and norepinephrine reuptake inhibitor. Oral MMEs are based on degree of mu-receptor agonist activity, but it is unknown if this drug is associated with overdose in the same dose-dependent manner as observed with medications that are solely mu receptor agonists.


# APPENDIX 8 SCHEDULE OF ASSESSMENTS - PHASE 1B MULTIPLE ASCENDING DOSE

**Table 4 Schedule of Assessments - Phase 1b - Multiple Ascending Dose** 

| | C 9 | ъ п | Treatment Period Follow-Up | | | | | | | | | | | Safety Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screena | Enroll | | | | | | 1 | | | ı | 1 | | | 1 | - |
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| GENERAL ASSESS | MENTS | | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| SLICC Criteria for<br>SLE | X | | | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>c</sup> | | X | | | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | | X | | X | X | X | X | X | | | | | |
| SAFETY ASSESSM | ENTS | ı | | | | | | | l | | l. | l. | | | l | 1 |
| Full physical exam | X | X | | | | | | | | | | | | | | |
| Chest x-ray <sup>d</sup> | X | | | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>e</sup> | X | X | | | X | | | X | | | | | | | | X |
| Injection site reaction assessment | | Xf | X | | X | | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | | X | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>g</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |


Table 4 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Tro | eatment | Period | Follow- | Up | | | | Safet | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | - | 11 | 12 | 13 |
| EFFICACY ASSESS | MENTS | | | | | | | | | • | | | | | | |
| BILAG-2004 Index | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLEDAI-2Kh | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| PGA of disease activity | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLICC/ACR<br>Damage Index | | X | | | | | | | | | X | | | | | |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| LABORATORY ASS | SESSMEN | TS | | | | | _ | | | | | | | | | |
| CD4+ count | X | X | | X | X | X | | X | | | X | | | | | |
| Clinical laboratory<br>assessments<br>(hematology and<br>clinical chemistry) <sup>i</sup> | X | X | | | X | X | X | X | X | X | X | | | X | X | X |
| Coomb's test direct | X | X | | | X | 21 | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | | X | X | X | 21 | X | 21 | 21 | X | | | 71 | 21 | 71 |
| Plasma CCI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Plasma CCI & | | X | | X | X | | X | X | | | X | | | | | |
| Whole blood for leukocyte immunophenotype | | X | | X | X | | X | X | | | X | | | | | |
| ADA <sup>k</sup> | | X | | X | X | | X | X | | | X | | | | | X |
| nAb <sup>l</sup> | | | | | | | | X | | | X | | | | | |
| pSTAT3 <sup>m</sup> | | X | | | X | X | X | X | | | | | | | | |
| CCI | | X | | X | | | | X | | | X | | | | | X |


Table 4 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Tre | eatment | Period | Follow- | Up | | | | Safet | y Follow | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| CCI | | X | | | | | | | | | | | | | | |
| CCI | X | X | | | X | | X | X | X | X | X | | | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> |
| CRP | X | 11 | | | 11 | | - 11 | X | 11 | 71 | 11 | | | - 11 | 11 | X |
| Serum pregnancy<br>test (women) | X | | | | | | | | | | | | | | | 11 |
| FSH<br>(postmenopausal<br>women) | X | | | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>o</sup> | | X | | | X | | X | X | X | X | X | | | | | X |
| TB test<br>(QuantiFERON-TB<br>Gold In-Tube) <sup>d</sup> | X | | | | | | | | | | | | | | | |
| Serology<br>(hepatitis B and C,<br>HIV-1/2<br>combination) | X | | | | | | | | | | | | | | | |
| Stool sample <sup>p</sup> | X | | | | | | | | | | | | | | | |
| Spot urine for protein/creatinine ratio | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | | X | | X | X | X | X | X | | | X | X | X |


 Table 4
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | | Safet | y Follow | v-Up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ | $(\pm 3)$ | (± 3) | $(\pm 3)$ | $(\pm 3)$ | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| PK Labs | | | | | | | | | | | | | | | | |
| Predose | | X | | | X | | X | X | X | X | X | | | | | |
| Predose PK<br>Window | | 60 m | | | ± 3 d | | ± 3 d | ± 3 d | ± 3 d | ± 3 d | ± 3 d | | | | | |
| Postdose | | Xq | X | X | Xq | | | | | | $X^q$ | X | X | X | X | X |
| Postdose PK<br>Window | | 4 h ±<br>30 m<br>8 h ±<br>45 m<br>24 h ±<br>60 m | ±1d | ±3 d | 4 h ±<br>30 m<br>8 h ±<br>45 m<br>24 h ±<br>60 m | | | | | | 4 h ±<br>30 m<br>8 h ±<br>45 m<br>24h ±<br>60 m | ± 3 d | ± 3 d | ± 3 d | ±3 d | ± 3 d |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; APL = antiphospholipid; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index;

CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; d = day; ECG = electrocardiogram;

; FSH = follicle stimulating hormone; h = hour; HR = heart rate; HIV = human immunodeficiency virus;

IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; m = minute; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SAE = serious adverse event; SC = subcutaneous; CC | SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; TB = tuberculosis; TDAR = T-cell dependent antigen response.

Screening assessments will be performed over more than 1 visit.

- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 4.6.1 for further details.
- <sup>c</sup> Randomization should occur after patient eligibility has been confirmed by central eligibility review.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- <sup>c</sup> ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed at 2 hours postdose.
- Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, 187, and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.


**Table 4** Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | Treatment Period Follow-Up | | | | | | | | | | Safety Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 7 15 30 44 60 90 120 150 180 187 195 | | | | | | | | 210 | 240 | 270 | | |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 1 | - | 11 | 12 | 13 |

- h SLEDAI-2K should be done before randomization and dosing on Day 0 as SLEDAI-2K < 6 is exclusionary.
- <sup>1</sup> Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be non-fasting.
- When clinically indicated for hemolytic anemia.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients, but only assayed (analyzed) if the patient had a positive ADA on Day 90.
- <sup>1</sup> nAb is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90.
- m Predose (trough) samples only.
- Antibodies and autoantibodies (CC) will not be analyzed during safety follow-up visits.
- <sup>o</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- P Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- Postdose samples will be collected at 4, 8, and 24 hours after study drug administration on Days 0, 30, and 180.


# APPENDIX 9 PROTOCOL SUMMARY OF CHANGES

The protocol summary of changes was moved to the end of the protocol for easier readability.

Significant changes are described in the table below. Changed text is displayed for the first major occurrence only. Deleted text is presented in strikethrough format, and added text is presented in bold format.

| Section | Description of Changes | Rationale |
|---|---|---|
| Global | Replace: | Administrative |
| | Protocol Date and Version: 23 January 2019; V5.0 | |
| | With: | |
| Global | Change: | Administrative |
| | Changed Version number from V5.0 (Amendment 4) to V6.0 (Amendment 5) and Version date from 23 January 2019 to 23 July 2019. | |
| Global | Made administrative and editorial (formatting, typographical, and grammatical) updates. | Administrative |
| CLINICAL<br>PROTOCOL | Replace: | Administrative |
| APPROVAL FORM | Name and Title | |
| | PPD , MD, FACR Vice President, Clinical Development Boston Pharmaceuticals | |
| | With: | |
| | Name and Title | |
| | PPD , PhD Senior Vice President | |
| | Clinical Development and Head of<br>Clinical Operations | |
| CLINICAL | Boston Pharmaceuticals Delete: | Administrative |
| PROTOCOL | | Administrative |
| APPROVAL FORM | Name and Title | |





| Section Protocol Date and Version | Description of Changes | Rationale |
|---|---|---|
| (sub-bullet 2) | | |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, MAD<br>Phase 1b, Exploratory | Replace: • CCI | CCI |
| Endpoints, Bullet 6 | With: | |
| Section 2.1, Study<br>Objectives and<br>Endpoints, Phase 1b<br>Multiple Ascending<br>Dose, Exploratory<br>Endpoints, Bullet 6 | • CCI | |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>Phase 2, Secondary<br>Endpoints, Bullet 1<br>(sub-bullet 3) | Replace: • The proportion of patients with: ○ a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210 | Protocol clarification |
| Section 2.2, Study<br>Objectives and<br>Endpoints, Phase 2<br>Proof of Concept,<br>Secondary Endpoints,<br>Bullet 1 (sub-bullet 3) | <ul> <li>With:</li> <li>The proportion of patients with:</li> <li>a sustained reduction from baseline of oral corticosteroid (CS) (≤ 7.5 mg/day and &lt; Day 0 dose) between Day 150 and Day 210</li> </ul> | |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>Phase 2, Secondary<br>Endpoints, Bullet 1<br>(sub-bullet 4) | Replace: • The proportion of patients with: • new BILAG A flare or > 1 BILAG B flares relative to baseline through Day 210 With: | Clarified to be<br>performed<br>against previous<br>visits, not only<br>baseline. |
| Section 2.2, Study<br>Objectives and<br>Endpoints, Phase 2<br>Proof of Concept,<br>Secondary Endpoints,<br>Bullet 1 (sub-bullet 4) | <ul> <li>The proportion of patients with:</li> <li>new or recurrent BILAG flares (≥ 1 qualifying BILAG A or &gt; 1 qualifying BILAG B) through Day 210</li> </ul> | |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>Phase 2, Secondary<br>Endpoints, Bullet 2 | Replace: Results and changes from baseline in: Swollen and tender joints ACR-28 With: | Clarified to<br>describe swollen<br>joint changes<br>from baseline. |


#### Section **Description of Changes** Rationale (sub-bullet 2) Results and changes from baseline in: Total number of swollen joints, tender joints, and Section 2.2, Study active joints (swelling and tenderness in the same Objectives and joint) in the ACR-28 joint count Endpoints Phase 2 Proof of Concept, Secondary Endpoints, Bullet 2 (sub-bullet 2) PROTOCOL Add: SUMMARY, Add endpoint to Objectives and Group mean percent reduction in CS administration measure overall Endpoints, POC from baseline Day 0 dose through Day 210 in patients CS reduction in Phase 2, Secondary patients receiving $\geq 7.5$ mg/day prednisone equivalent at Day 0 Endpoints, Bullet 4 receiving CS at baseline. Section 2.2, Study Objectives and Endpoints, Phase 2 Proof of Concept, Secondary Endpoints, Bullet 4 PROTOCOL Replace: SUMMARY, Clarified this is Objectives and for the time to Time to BILAG A flare or > 1 BILAG B flare compared to Endpoints, POC first flare and baseline through Day 210 Phase 2, Secondary allowed for new Endpoints, Bullet 7 or recurrent With: BILAG flare to Section 2.2, Study allow for Time to first BILAG flare (≥ 1 new or recurrent Objectives and improvement **BILAG A** or > 1 new or recurrent BILAG B) relative to Endpoints, Phase 2 and subsequent baseline through Day 210 Proof of Concept, worsening. Secondary Endpoints, Bullet 7 PROTOCOL Delete: SUMMARY, Objectives and Endpoints, POC Phase 2, Exploratory **Endpoints** (Pharmacodynamic) Section 2.2, Study Objectives and Endpoints, Phase 2 Proof of Concept, **Exploratory Endpoints** (Pharmacodynamic)


#### Section

## **Description of Changes**

#### Rationale

Protocol

clarification.

PROTOCOL SUMMARY, Study Design, Paragraph 5 Replace:

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 60. Tapering of steroids during the course of the study will be highly encouraged and should be evaluated at the protocol permitted visits (Day 0 through Day 60 and Day 120 through Day 150). Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant due to the endpoint evaluations occurring at Day 120 and Day 210.

With:

A maximum stable (for at least 6 weeks prior to Day 0) daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study. One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 120. Tapering of steroids during the course of the study will be highly encouraged and should be evaluated during the protocol-allowed tapering windows (Day 0 through Day 150) with the target of achieving a CS daily dose of ≤ 7.5 mg and < Day 0 dose between Day 150 and Day 210. Between Day 150 and Day 210, oral CS doses must be held constant due to the Day 210 endpoint evaluations.

PROTOCOL SUMMARY, Main Criteria for Inclusion and Exclusion, Inclusion Criteria, criteria 4, c

Section 4.4, Inclusion Criteria, criteria 4, c

PROTOCOL SUMMARY, Main Criteria for Inclusion and Exclusion, Inclusion Criteria, criteria 5 Delete:

c. CCl levels below normal as determined by the central lab

Allowing patients to enroll on low compliment alone is not specific enough for SLE.

#### Replace:

- 5. At screening, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - Points from lupus headache and organic brain syndrome will also be excluded

With:

5. At screening, the **total** SLEDAI-2K **score** must be  $\geq$  **8**, including

To ensure patients with Moderate to Severe active disease are enrolled.


#### Section Description of Changes

#### Rationale

points from at least 1 of the following clinical components:

a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

# PROTOCOL SUMMARY, Main

Criteria for Inclusion and Exclusion, Inclusion Criteria, criteria 6

Section 4.4, Inclusion Criteria, criteria 6

Replace:

- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - Points from lupus headache and organic brain syndrome will also be excluded

With:

- 6. A clinical SLEDAI-2K score of ≥ 6 at screening at Day 0. Clinical SLEDAI-2K score is defined as follows:
  - a. Contains points from arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, or vasculitis
  - b. Excludes parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

PROTOCOL SUMMARY, Main

Criteria for Inclusion and Exclusion, Inclusion Criteria, criteria 7 Replace:

- 7. Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined in the protocol Section 4.4

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

With:

7. Patients must have at least 1 **qualifying** A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the

To ensure patients with Moderate to Severe active disease are enrolled.

To ensure patients with Moderate to Severe active disease are enrolled.

Clarification of active joint term.


#### Section

# **Description of Changes**

Rationale

central data reviewer:

- a. BILAG A or B score in the mucocutaneous body system. If a BILAG B score is due to BILAG number 6, mild skin eruption, the CLASI activity score including erythema and scale/hypertrophy must be ≥ 3 excluding points from mucosal ulcers and alopecia.
- b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined in the protocol Section 4.4

Note: Hips, shoulders, back, neck, and temporomandibular joints do not count towards the total number of joints with active synovitis.

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in **at least 1** other body system for a total of **2** "B" BILAG body system scores.

PROTOCOL SUMMARY, Main Criteria for Inclusion and Exclusion, Inclusion Criteria,

Section 4.4, Inclusion Criteria, criteria 8

criteria 8

#### Replace:

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization)

#### With:

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to **Day 0**) of the following permitted steroid-sparing agents:
    - Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. If AZA, myocophenolate mofetil, mycophenolic acid, hydroxychloroquine, or MTX were discontinued prior to screening, the washout period must be ≥ 12 weeks.
  - c. Corticosteroids (prednisone or prednisone-equivalent) at a stable dose of up to 30 mg/day for at least 6 weeks prior to Day 0 (see APPENDIX 3)
    - i. For patients whose only SLE treatment is CSs, the stable CS dose must be  $\geq 10$  mg/day for at least 6 weeks prior to Day 0 and no more than 30 mg/day at the time of randomization.
    - ii. Topical steroids may be used, but the dose must be stable for at least 6 weeks prior to Day 0. PRN topical

A stable dose is needed 8 weeks prior to Day 0; it is not necessary to be longer.

Removed the tapering requirement prior to randomization, determined not to be required.

To ensure patients with Moderate to Severe active disease are enrolled.


| Section Section | Description of Changes | Rationale |
|---|---|---|
| | steroids are not permitted. | |
| PROTOCOL<br>SUMMARY, Main | Add: | To clarify that sponsor or |
| Criteria for Inclusion<br>and Exclusion,<br>Exclusion Criteria<br>criterion 7, 23, and 27 | 7. Concomitant illness that, in the opinion of the investigator <b>or the sponsor or their designee</b> , is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary | designee can<br>determine a<br>patient is not<br>eligible. |
| Section 4.5, Exclusion<br>Criteria, criterion 7, | 23. Any other laboratory test results that, in the opinion of the Investigator <b>or the sponsor or sponsor's designee</b> , might place a patient at unacceptable risk for participating in this study | |
| 23, and 27 | 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, <b>sponsor or sponsor's designee</b> , would make the patient inappropriate for entry into this study | |
| PROTOCOL<br>SUMMARY, Main | Replace: | Reduced based on safety data |
| Criteria for Inclusion | 15. CD4+ count < 350/μL at screening | from MAD |
| and Exclusion, Exclusion Criteria | With: | portion of the study. |
| criterion 15 | 15. CD4+ count < <b>150</b> /μL at screening | |
| Section 4.5, Exclusion<br>Criteria, criterion 15 | | |
| PROTOCOL | Replace: | Total bilirubin is |
| SUMMARY, Main<br>Criteria for Inclusion<br>and Exclusion, | 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome) | tested at screening, but direct bilirubin |
| Exclusion Criteria criterion 22 | With: | is only tested when there is |
| Section 4.5, Exclusion<br>Criteria, criterion 22 | 22. <b>Total</b> bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome) | potential liver injury. |
| PROTOCOL | Add: | Opioid will |
| SUMMARY, Main<br>Criteria for Inclusion<br>and Exclusion,<br>Exclusion Criteria<br>criterion 33 | 33. Currently taking a total daily dose of > 30 mg morphine or morphine equivalent (see Appendix 7) | mask SLE<br>symptoms. |
| Section 4.5, Exclusion<br>Criteria, criterion 33 | | |
| PROTOCOL<br>SUMMARY, Main | Add: | Added restriction due |
| Criteria for Inclusion and Exclusion, | 34. Body mass index (BMI) $\geq$ 40.0 | to increased co-morbidities |


| Section Section | Description of Changes | Rationale |
|---|---|---|
| Exclusion Criteria criterion 34 | | in patients with<br>high BMI that<br>will hinder SLE |
| Section 4.5, Exclusion<br>Criteria, criterion 34 | | Assessments. |
| LIST OF<br>ABBREVIATIONS | Add: | Terms added to protocol |
| | ADL activities of daily living | amendment. |
| | BMI body mass index | |
| | NSAID nonsteroidal anti-inflammatory drug | |
| Section 3.1.2.1,<br>BOS161721 POC | Replace: | Protocol clarification. |
| Dose Selection and<br>Justification,<br>Paragraph 5 | The 120 mg dose will be communicated to site investigators participating in the POC Phase 2 portion, and to Institutional Review Boards (IRBs) and the Independent Ethics Committee (IEC). | |
| | With: | |
| | The 120 mg dose <b>was</b> communicated to site investigators participating in the POC Phase 2 portion, and to Institutional Review Boards (IRBs) and the Independent Ethics Committee (IEC). | |
| Section 3.1.2.2, POC<br>Study Design, | Replace: | Protocol clarification. |
| Paragraph 2 | As in the MAD part of the study, each patient in the POC portion may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Section 3.4). | ciarmeanon. |
| | With: | |
| | As in the MAD part of the study, each patient in the POC portion may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments ( <b>Table 1 and Table 4</b> ). | |
| Section 3.4, Schedule of Assessments, Table 1 | Delete: | Since Phase 1b<br>MAD has<br>completed, the<br>Schedule of<br>Assessments for<br>Phase 1b MAD<br>was moved to<br>the Appendix. |


#### Section Description of Changes

Rationale

| _ | Screen | Enrol<br>lo | | | | Tee | aimeni | Period | Follow | Upra | | | | | Follow | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 0 | | - Ro | | | | | | | | | | | | | | |
| David | -28· | 4a | 24<br>(49)o | 35¶<br>(±/3)o | 30¶<br>(4/3)o | 44¶<br>(4/8)o | 60¶<br>(+03)o | 905<br>(6/3) | 120¶<br>(±3)c | 350¶<br>(±'3)c | 180¶<br>(4/0)o | 187¶<br>(±03)o | 1955 | 210¶<br>(±03)u | 248¶<br>(±/3)o | 2709<br>(±/3): |
| Visit/Numbero | la | 20 | -0 | 30 | -4a | ≨a. | 6a | 7a | \$o | 9o | 10a | -0 | -0 | 11a | 12a | 130 |
| GENERAL ASSESS | MENTS | | | | | | | | | | | | | | | |
| · Informed-consent: | Xo. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Inclusion Exclusion | | | 0 | | | | | | | | | ō | 0 | | | |
| criteria: | Xo. | 0 | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | | | 0 | 0 | .0 |
| •Medical-history: | Xo. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| •Demographics⊃ | Xo. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| SLICC-Criteria for<br>SLE-0 | Xo. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Concomitant<br>medication <sup>b</sup> | Xo. | Xo. | Xo. | Χo | Xo. | Xo. | Χo | Xo. | Χo | Xo. | Xo. | Xo. | Xo. | Xο | Xo. | No. |
| •Randomization* | 0 | No | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| *B08161221-or | _ | | | - | _ | _ | - | _ | - | - | - | | | _ | - | _ |
| placebo-dosing © | | Xo. | | | Xo. | | Xo. | Xo. | Xo | Xo. | Xo. | | " | | | 0 |
| SAFETY-ASSESSM | ENTSo | | _ | _ | | | | | | | | | | | _ | |
| Full-physical-exam? | Xo | Xo | 0 | 0 | 0 | | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 |
| • Chectos-ray <sup>4</sup> 0 | Xo. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| C SSRS: | Xo. | Xo. | 0 | 0 | 0 | 0 | 0 | Xo. | 0 | 0 | Xο | 0 | 0 | 0 | 0 | .0 |
| ·AEs and SAEso | 0 | Xo | Xo | Xo | Xo | Xo | Xo | Xo | Xo | Xο | Xo | Xo | Xo | Xo | Xo | Xo |
| •12 lead ECG*: | Xo. | Xo | 0 | 0 | Xo | 0 | 0 | Xo | 0 | 0 | 0 | 0 | 0 | 0 | 0 | Xo |
| *laiection-site | | | | | | | | | | | | | | | | |
| reaction-assessment* | 0 | X <sup>i</sup> o | Xo | 0 | Xo | 0 | Xo | Xo | Xo | Xo | Xo | Xo | Xo | Xo | Xo | Xo |
| Targeted physical examination | | | 0 | Хo | Хo | Xo | Xo | Xo | Xo | Xo. | Xo | 0 | 0 | Xo | Xo. | Xo |
| Vital eigns (BP, HR, | _ | | 0 | - 1 | | | - 11 | | | | | 0 | 0 | | - 11 | |
| and temperature)F | Xo | Xo | | Xo | Xo | Xo | Xo | Xo | Xo | Xo | Xo | | | Xo | Xo | Xo |

| 0 | Screen<br>to | Enrol<br>lo | | | | Tre | atment | Period: | Follow | Upro | | | | Safet | Follow | Upo |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dayso | -28-<br>tola | ₩a | 34<br>(4/8)o | 15¶<br>(4/5)a | 30¶<br>(4/3)¤ | 44¶<br>(#3)a | 60¶<br>(4/0)o | 90¶<br>(4/3)o | 120¶<br>(4/3)c | 150¶<br>(4/3)c | 150¶<br>(4/3)o | 1875<br>(4/3)o | 195¶<br>(4/3)c | 210¶<br>(4/3)a | 240¶<br>(#/8)c | 270¶<br>(4/3)c |
| VisitNumber: | lo | 2a | -0 | 3o | 40 | \$a | 6a | <b>3</b> a | S <sub>O</sub> | 9a | 100 | -0 | -0 | 11a | 12a | 13a |
| EFFICACY-ASSESS | MENTS: | | | | | | | | | | | | | | | |
| BILAG 2004 Index | Xo. | Xo. | 0 | 0 | Xo. | 0 | Xo. | Xo. | Xo. | Xo. | Xo. | 0 | 0 | Xο | Xo. | Xo. |
| SLEDAI 2Kin | Xo. | Xo. | 0 | 0 | Χo | 0 | No. | Xo. | Xo. | Xo. | Xo. | 0 | 0 | Χo | Xo. | Xo. |
| PGA-of-disease | | | 0 | | | | | | | | | 0 | 0 | | | |
| activityo | Xo. | Xo. | | 0 | Xo. | 0 | Xo. | Xo. | Xo. | Xo. | Xo. | | | Xo. | Xo. | Xo. |
| ACR 28 joint count | Xo. | Xo. | 0 | 0 | Χo | 0 | Xo. | Xo. | Xo. | Xo. | Xo. | 0 | 0 | Χo | Xo. | Xo. |
| -CLASIo | Xo. | Xο | 0 | 0 | Χo | 0 | Xo. | Xo. | Xo. | Xo. | Xo. | 0 | 0 | Xo. | Xo. | Xo. |
| CCI | 0 | Xo | 0 | 0 | Χo | 0 | Χo | Χo | Xo | Xo | Χo | 0 | 0 | Χo | Xo | Xo |
| SLICC/ACR | | | 0 | | | | | | | | | 0 | 0 | | | |
| Damage-Index≎ | 0 | Xo | | 0 | 0 | .0 | 0 | 0 | 0 | 0 | Xo | | | 0 | 0 | 0 |
| CCI | 0 | Χo | 0 | | Χo | 0 | Жo | Χo | Χo | Xo | Χo | 0 | 0 | Жo | Жo | Xo |
| LABORATORY AS | SESSME: | CSTA | | | | | | | | | | | | | | |
| CD4+-count0 | Xo. | Xo. | 0 | Χo | Χo | Xo. | 0 | Xo. | 0 | 0 | Xο | 0 | 0 | 0 | 0 | 0 |
| Clinical laboratory | | | 0 | | | | | | | | | 0 | 0 | | | |
| accessments: | | | | | | | | | | | | | | | | |
| (hematology-and | | | | | | | | | | l l | | | | | | |
| olinical obemistry) <sup>j</sup> □ | Xo. | Xο | | 0 | Xο | Xο | Xο | Xο | Xο | Xo. | Xο | _ | | Xο | Xο | Xo |
| Coomb's test-direction | Xo. | Xo. | 0 | 0 | Xο | 0 | X0 | Xo. | Xο | Xo. | Xο | 0 | ٥ | Xo. | Xo. | Xo. |
| Total-IgG-and-IgM o | Xo. | Xο | 0 | Xο | Xo. | Xo. | 0 | Xo. | 0 | ٥ | Xο | 0 | 0 | 0 | 0 | 0 |
| CCI | Xo | X.o | 0 | 0 | Xο | 0 | X.o | Xo | Χo | Xo | Xο | 0 | 0 | Xo | Xo | Xo |
| CCI | 0 | Xο | ۰ | Χo | Xο | 0 | Χo | Χo | 0 | 0 | Xο | 0 | 0 | 0 | 0 | 0 |
| Whole-blood-for- | | | 0 | | | | | | | | | 0 | 0 | | | |
| ieukocyte<br>immunophenotype: | 0 | Χo | | Xο | Xo | 0 | Xo | Xo | о | 0 | Xο | | | 0 | 0 | 0 |
| ADA** | 0 | Xo. | 0 | Xo. | Xo. | 0 | No. | Xo. | 0 | 0 | Xo. | 0 | 0 | 0 | 0 | Xo. |
| nAli/o | 0 | 0 | 0 | 0 | 0 | 0 | 0 | Χo | 0 | 0 | Xo. | 0 | 0 | 0 | 0 | 0 |
| pSTAT2 <sup>20</sup> 0 | 0 | Xo. | 0 | 0 | Χo | Xo | Xo | Xo | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

| а | Screen | Enrol<br>lo | | | | Tre | atment | Period | Follow | Upm | | | | Safet | y-Follow | -Upa |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dayeo | -28-<br>to-lo | Øg. | 24<br>(49): | 15¶<br>(±13)o | 30¶<br>(#3)a | 44¶<br>(4/3)o | 69¶<br>(+9)o | 90¶<br>(+33)c | 120¶<br>(±/3)o | 150¶<br>(±33)o | 180¶<br>(±/3)o | 1875<br>(+03)c | 195¶<br>(±/3)o | 210¶<br>(±/3)α | 246¶<br>(±93)o | 270¶<br>(±'3): |
| Visit/Numbero | la | 20 | -0 | 3o | 40 | \$a | 6a | 30 | Sc. | 90 | 10a | -0 | -0 | 11 <sub>0</sub> | 120 | 13 <sub>0</sub> |
| CCI | 0 | Xo | 0 | X: | 0 | 0 | 0 | Xo. | 0 | 0 | Xo. | 0 | 0 | 0 | 0 | No. |
| | | Xo | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| CCI | Xo. | Xo. | 0 | _ | Xo. | | Xo | Xo. | Xo. | Xo. | Xo | 0 | 0 | XPo | XPo | X4o |
| CRPo | Xo | 0 | 0 | 0 | 0 | 0 | 0 | Xo | 0 | 0 | 0 | 0 | 0 | 0 | 0 | Xo. |
| Serum-precnancy | 20 | | 0 | 0 | 0 | - 0 | 0 | - A-0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | A0 |
| test-(women): | X- | | ۰ ا | | | | 0 | | | | | | | 0 | | |
| FSH | - | | 0 | | | | | | | | | 0 | 0 | | | |
| (postmenopausal-<br>women)© | Xo. | | | ٥ | ٥ | | 0 | ٥ | 0 | ٥ | ٥ | | | ٥ | ٥ | 0 |
| Urine pregnancy<br>test (women) <sup>2</sup> 0 | | Χo | 0 | 0 | Χo | | Χo | Χo | Χo | Χo | Xο | 0 | 0 | 0 | 8 | Χo |
| TB-test | | | 0 | | | | | | | | | 0 | 0 | | | |
| (QuantiFERON TB<br>Gold In Tube)40 | X0 | ۰ | | | 0 | | 0 | | 0 | | | | | 0 | | 0 |
| Serology (hepatitis<br>B and C. HIV 1/2 | | | ٥ | | | | | | | | | ٥ | 0 | | | |
| combination): | Xo | 0 | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | | | 0 | 0 | 0 |
| Stool-cample <sup>p</sup> | Xo | 0 | 0 | 0 | ٥ | 0 | 0 | Ö | 0 | 0 | 0 | ٥ | 0 | ٥ | Ö | 0 |
| Spot-unine-for protein creatinine | | | 0 | | | | | | | | | 0 | 0 | | | |
| ratio | X0 | Xo. | | 0 | Xo. | 0 | Xo. | Xo. | X0 | Xο | Xο | | | Xo. | Xο | Xo. |
| Urinalysis | Xo | Xo | 0 | 0 | Xo | 0 | Xo | Xo | Xo | Xo | Xo | 0 | 0 | Xo | Xo | Xo |

| | Screen* | Enroll | | | | In | eatment | Period | Follow | Up | | | | Safet | y Follow | -Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dave | -28<br>to 1 | a | (4-1) | 15<br>(a-3) | 30<br>(±3) | 44<br>(a-3) | 60<br>(a.3) | 90<br>(a.3) | 120<br>(±-3) | 150<br>(±-3) | 180<br>(±-3) | 187<br>(a-3) | 195<br>(±-3) | 210<br>(±3) | 240<br>(a-3) | 270<br>(a.3) |
| Visit Number | 1 | 2 | - | 3 | 4 | | 6 | 2 | 8 | 9 | 10 | - | - | 11 | 12 | 13 |
| PK Labs | | | _ | | | | | | | | | | _ | | | |
| Predose | | x | | | x | | x | X | X | X | x | | | | | |
| Predoce PK<br>Wandow | | 60m | | | +34 | | +34 | +34 | +34 | -34 | +34 | | | | | |
| Postdose | | X9 | x | х | 23 | | | | | | 309 | x | x | X | X | X |
| Postdore PK<br>Window | | 30m<br>8h =<br>15m<br>21h =<br>50m | <u>+14</u> | <u>- 34</u> | 20m.<br>80m.<br>45m.<br>210m. | | | | | | 4h-a<br>30m<br>8h-a<br>45m<br>24h-a<br>60m | <del>+ 3d</del> | <u>-34</u> | <u>+34</u> | <del>- id</del> | ±-34 |
| Abbreviations: AC<br>Lupus Assessment<br>CRP = C reactive o<br>CC<br>InG = immunoclob | Group; BP =<br>rotein: C SSI | blood pred<br>LS = Colu | mure; C<br>mbia St<br>FSH = 1 | = comp<br>sicide Se<br>follicle s | lement; (<br>everity Ra<br>timulatio | D4 = c<br>sting Scal<br>g hormor | iuster of<br>ie; d = d<br>ne; h = h | differen<br>sy: ECG<br>our: HR | melectr<br>= heart | CLAS<br>coardio<br>rate; HI | ram: | C I | eus Are<br>nodelies | escy viru | erity Ind | law) |


#### Section

#### **Description of Changes**

Rationale



Section 3.4, Schedule of Assessments, Table 1 footnote "c"

#### Replace:

Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0.

With:

<sup>c</sup> Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the dose must be stable for at least 6 weeks prior to Day 0.

Section 3.4, Schedule of Assessments, Table 1 footnote "n"

#### Replace:

Only CCl collected during safety follow-up visits.

With:

not be analyzed during safety follow-up visits.

Section 3.4, Schedule of Assessments, Table 1, Whole blood leukocyte immunophenotype row

#### Delete:

| • p | Screen | Enrolla | | | T | reatmen | t-Period: | Follow-u | pπ | | | Safet | w-Upa | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15¶ | 30¶ | 60¶ | 90¶ | 120¶ | 150¶ | 180¶ | 1875¶ | 195b¶ | 210¶ | 240¶ | 270¶ |
| ■Days¤ | to-l¤ | 0α | (±°3)¤ | (±3)¤ | (±3)α | (±3)a | (±3)a | (±3)¤ | (±%)¤ | (±3)¤ | (±°3)α | (±°3)∷ | (±%)¤ | (±%)¤ |
| • Visit Numbera | lα | <b>2</b> α | <b>3</b> ⊠ | 4¤ | 5¤ | <b>6</b> ¤ | 7¤ | <b>8</b> ¤ | 9≅ | à | ¤ | 10¤ | 11¤ | 12¤ |
| <ul> <li>LABORATORY-ASSESSMENT</li> </ul> | S≎ | | | | | | | | | | | | | |
| Whole blood for leukocyte | | | | | | | | | | a | 0 | | | |
| immunophenotype <sup>□</sup> | Ö | ¥ο | Xο | Xο | a | Xο | 0 | 0 | ¥ο | | | ۵ | ۵ | ٥ |

Section 4.3, Patient Screening

Replace:

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Section 3.4]) for this

Protocol clarification.

Correcting error in protocol.

This data is no longer necessary; the MAD data collected has been sufficient.

Protocol clarification.


#### Section

#### **Description of Changes**

Rationale

To ensure

patients with

Moderate to

disease are enrolled.

Severe active

study must be performed between Day -28 and Day -1.

With:

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Table 1 and Table 4]) for this study must be performed between Day -28 and Day -1

# Section 4.4, Inclusion Criteria, criteria 5

#### Replace:

- 5. At screening, the SLE Disease Activity Index 2000 (SLEDAI-2K) must be ≥ 6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - Points from lupus headache and organic brain syndrome will also be excluded

#### With:

- 5. At screening, the **total** SLEDAI-2K **score** must be  $\geq$  **8**, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis

Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.

# Section 4.4, Inclusion Criteria, criteria 7

#### Replace:

- 7. Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis in ≥ 2 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living that has been present on several days cumulatively over the past 30 days, including at the time of the screening visit. See

To ensure patients with Moderate to Severe active

disease are enrolled.

Clarification of active joint term.


#### Section Description of Changes

Rationale

APPENDIX 5 for additional detailed specifications.

- Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):
  - Ambulation, toileting, grooming- including bathing and dressing; feeding oneself
- ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in ≥ 1 joint, (observed or throughout history), with some loss of functional range of movements manifested by effects on instrumental ADLs such as:
  - Cooking, driving, using the telephone or computer, shopping, cleaning, etc., and has been present on several days over the last 30 days, and is present at the time of the screening visit

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

#### With:

- 7. Patients must have at least 1 qualifying A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system. If a BILAG B score is due to BILAG number 6, mild skin eruption, the CLASI activity score must be ≥ 3 excluding points from mucosal ulcers and alopecia.
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - i. "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis defined by BOTH swelling and tenderness in ≥ 6 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living (ADLs) that has been present on several days (> 4 days).cumulatively over the past 30 days, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
      - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):
        - Ambulation, toileting, grooming- including bathing and dressing; feeding oneself
    - ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis defined by BOTH swelling and tenderness in ≥ 3 joints, (observed or through patient history), with some loss of functional range


#### Section Description of Changes

Rationale

of movements manifested by effects on instrumental ADLs such as:

• Cooking, driving, using the telephone or computer, shopping, cleaning, etc., and has been present on several days over the last 30 days, and is present at the time of the screening visit

Note: Hips, shoulders, back, neck, and temporomandibular joints do not count towards the total number of joints with active synovitis.

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in **at least 1** other body system for a total of 2 "B" BILAG body system scores.

Section 4.6, Concomitant Medications Add:

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Patients should stay on stable regimen (not PRN) of other concomitant medications for the treatment of SLE (eg, analgesics, nonsteroidal anti-inflammatory drugs [NSAIDs], statins, ACE inhibitors/ARBs and other antihypertensive drugs), unless changes in these treatments are clinically indicated. Patients should refrain from Tylenol, NSAIDs, and any pain medications including tramadol and other opiates for at least 12 hours before each visit, with the exception of the Screening Visit.

Use of any other drugs for non-SLE conditions, including over-the-counter medications and herbal preparations, should remain stable unless change or addition is clinically necessary. Discussion with the medical monitor prior to initiation of new medication is strongly recommended. Any concomitant therapies must be recorded on the eCRF. Prior and concomitant medication use will be recorded for the 30 days prior to screening until the last follow-up visit. In addition, historical treatment for SLE (including immunosuppressant, anti-malarial, corticosteroid, and/or biologic agent **including investigational agents**) will be recorded for the 48 weeks prior to screening in the eCRF.

Section 4.6.1, Corticosteroid

Replace:

#### 4.6.1 Oral Corticosteroid Dose

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day).

Protocol clarification.

Protocol text further clarified to include investigational agents.

Added further clarity to section regarding tapering and allowed burst Removed the restrictions of max burst dose and extended protocol allowed burst window to assist sites in managing their patients SLE. Text modified to


BOS161721 Boston Pharmaceuticals, Inc.


#### Section Descri

#### **Description of Changes**

Tapering of steroids during the course of the study will be highly encouraged and should be evaluated at the protocol permitted visits (Day 0 through Day 60 and Day 120 through Day 150). Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant due to the endpoint evaluations occurring at Day 120 and Day 210.

- Once a patient has received the first dose of study drug (after Day 0), prednisone (or prednisone equivalent) dose is highly encouraged to continue tapering down as appropriate. The investigator should evaluate the prednisone dose at each visit and make the decision, within the protocol allowed windows.
  - Exception: Between Day 60 and Day 120, and between Day 150 and Day 210 (ie, within 60 days of primary and secondary endpoint assessments), oral CS doses must be held constant.

After Day 0 (first dose of study drug), a maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed between Day 0 and Day 60, according to the following:

- The oral CS dose is allowed to increase to ≤ 40 mg/day of prednisone or equivalent, which must be tapered down to ≤ 10 mg/day within 2 weeks of initiation of the "burst"
  - Alternatively, a single intramuscular (IM) dose of methylprednisolone (40 mg or equivalent) is permitted
  - No increase of oral CS above baseline is permitted beyond Day 60

Treatment with inhalational CS therapy (eg, for asthma), or by any other route, but systemic administration, is allowed.

Treatment with intra-articular or intravenous CS is prohibited during the course of the study.

#### With:

#### 4.6.1 Corticosteroid

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study. For patients whose only SLE treatment is steroids, their stable steroid dose must be at least 10 mg/day and no more than 30 mg/day for a minimum of 6 weeks at time of randomization on Day 0.

Topical steroids may be used, but the dose must be stable for at

Rationale

ensure patients with Moderate to Severe active disease are enrolled.

Further clarification of protocol intention.


#### Section Description of Changes

Rationale

least 6 weeks prior to Day 0, and be maintained at a constant dose throughout the study duration until the rashes resolve. PRN topical steroids are not permitted.

Once the patient has received the first dose of study drug (Day 0), tapering of oral steroids will be highly encouraged and should be continually evaluated during the protocol-allowed tapering windows (Day 0 through Day 150) with the target of achieving a CS daily dose of < 7.5 mg and < Day 0 dose between Day 150 and Day 210.

Between Day 150 and Day 210 (ie, within 60 days of primary endpoint assessments), oral CS doses must be held constant.

#### CS Burst for SLE-related Indications

After Day 0 (first dose of study drug), a maximum of 1 oral CS "burst" equivalent to  $\leq$  40 mg/day prednisone for increased SLE disease activity will be allowed between Day 0 and Day 120, which must be tapered down to the baseline (Day 0) CS dose or lower within 14 days of initiation of the "burst." Any "burst" continuing after Day 120 or occurring after Day 120 is considered a protocol deviation.

 Alternatively, a single intramuscular (IM) dose of methylprednisolone (<40 mg) is permitted during this period.

#### CS Burst for Non-SLE-related Indications

A single treatment of oral prednisone equivalent of  $\leq$  40 mg/day for 14 days is permitted for a non-SLE indication, though it must be completed prior to Day 120. No long acting steroid injections are permitted.

Note: Treatment with inhaled CS are allowed for the treatment of non-SLE-related indications only (eg, for asthma).

Any other increase from baseline of CS dose or systemic use of CS of any kind (including intra-articular and intravenous administration) are not permitted from Day 0 through Day 210 and will result in the patient being considered a treatment failure. There is no restriction of CS usage after Day 210.

Section 4.6.2, Other Prohibited and/or Restricted Treatments, Paragraph 1 Replace:

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in APPENDIX 4. Medications taken within 30 days prior to screening must be recorded on the eCRF.

Protocol clarification.


#### Section Description of Changes Rationale

With:

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in APPENDIX 4. **All medications** taken within 30 days prior to screening must be recorded on the eCRF.

Section 4.6.2, Other Prohibited and/or Restricted Treatments, Item 2 Delete:

2. Patients who have received treatment with anti-CD20 monoclonal antibodies within 24 weeks of screening; recovery of B cells (CD19+) must be documented (record absolute number of CD19+B cells)

Protocol text removed as it was no longer necessary.

Section 4.7.2, Contraception, Paragraph 4 Replace:

At a minimum, patients must agree to the use of 1 method of highly effective contraception from the following:

To ensure patients have appropriate contraception during the study.

With:

Patients must agree to either complete abstinence, defined as a complete avoidance of heterosexual activity, or the use of 2 methods of highly effective contraception from the following:

Section 4.7.2, Contraception, Paragraph 4, Bullet 4 and 5 Replace:

Protocol clarification.

- Vasectomy
- Complete abstinence, defined as complete avoidance of heterosexual intercourse, is an acceptable form of contraception.
   Women who are abstinent while participating in the study must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the patient chooses to forego complete abstinence.

With:

Vasectomy

**Note:** Women who are abstinent while participating in the study must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the patient chooses to forego complete abstinence.

Section 5.1, Screening, Paragraph 5 Replace:

Protocol clarification.

Screening procedures are listed in the Schedule of Assessments (Section 3.4), and details are provided in Section 6.

With:

Screening procedures are listed in the Schedule of Assessments


| Section | Description of Changes | Rationale |
|---|---|---|
| | (Table 1 and Table 4), and details are provided in Section 6. | |
| Section 5.2,<br>Enrollment/<br>Randomization and<br>Day 0 Treatment,<br>Paragraph 1 | Add: Randomization should occur after patient eligibility for enrollment has been confirmed by the central eligibility review. The central eligibility review team has the final decision on patient eligibility and can decide the patient is not eligible for the study based on their review of the eligibility packet. | To provide further clarification that the central eligibility review team can deem a patient in-eligible for randomization even if all entrance criteria are met. |
| Section 5.2,<br>Enrollment/ | Add: | No longer |
| Randomization and | • Laboratory evaluations (fasting): | necessary in POC portion of |
| Day 0 Treatment,<br>bullet 3, sub-bullet 3 | o CD4+ count, total IgG and IgM levels, plasma CCl plasma CCl and and CCl who whole blood for leukocyte immunophenotype (leukocyte immunophenotype for MAD patients only) | the study. MAD data collected has been sufficient. |
| Section 5.2,<br>Enrollment/ | Replace: | Protocol clarification. |
| Randomization and | • Laboratory evaluations (non-fasting): | orar mounton. |
| Day 0 Treatment,<br>bullet 3, sub-bullet 9 | <ul> <li>See Table 1 and Table 2 for details of PK sampling in the<br/>MAD and POC portions</li> </ul> | |
| | With: | |
| | • Laboratory evaluations (non-fasting): | |
| | <ul> <li>See Table 4 and Table 1 for details of PK sampling in the<br/>MAD and POC portions</li> </ul> | |
| Section 5.2,<br>Enrollment/ | Replace: | Protocol clarification. |
| Randomization and Day 0 Treatment, Paragraph 4 | Procedures on Day 0 are listed in the Schedule of Assessments (Section 3.4), and details are provided in Section 6. | Claimeanon. |
| r aragrapii 4 | With: | |
| | Procedures on Day 0 are listed in the Schedule of Assessments ( <b>Table 1</b> and <b>Table 4</b> ), and details are provided in Section 6. | |
| Section 5.3, | Replace: | Protocol |
| Treatment<br>Period/Follow-Up<br>Visits, Pararaph 1 and<br>bullet 17 | The following procedures will be performed as indicated in the Schedule of Assessments (Table 1 and Table 2). See Schedule of Assessment tables for allowable windows for each visit. | clarification. |
| | • See Table 1 and Table 2 for details of PK sampling in the MAD | |


#### Section Desc

#### Description of Changes Rationale

and POC studies, respectively

With:

The following procedures will be performed as indicated in the Schedule of Assessments (**Table 1** and **Table 4**). See Schedule of Assessment tables for allowable windows for each visit.

 See Table 4 and Table 1 for details of PK sampling in the MAD and POC studies, respectively

#### Section 5.3,

Treatment
Period/Follow-Up
Visits, bullet 20

#### Replace:

Plasma CCl & CCl , ADA, and whole blood for leukocyte immunophenotype

#### With:

 Plasma CC and CC , ADA, and whole blood for leukocyte immunophenotype (leukocyte immunophenotype for MAD patients only)

Section 5.4, Safety Follow-Up Visits, Paragraph 1 and bullet 18

#### Replace:

Safety follow-up visits will take place at Days 210, 240, and 270. These visits will include the following assessments as indicated in the Schedule of Assessments (Table 1 and Table 2):

 See Table 1 and Table 2 for details of PK sampling in the MAD and POC portions, respectively

#### Replace:

Safety follow-up visits will take place at Days 210, 240, and 270. These visits will include the following assessments as indicated in the Schedule of Assessments (**Table 1** and **Table 4**):

 See Table 4 and Table 1 for details of PK sampling in the MAD and POC portions, respectively

#### Section 6.2.1, Laboratory Assessments, Paragraph 1

#### Replace:

Laboratory tests will be performed at times defined in the Schedule of Assessments (Section 3.4). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

#### With:

Laboratory tests will be performed at times defined in the Schedule of Assessments (**Table 1 and Table 4**). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived

No longer necessary for POC portion of study. MAD data collected has been sufficient.

Protocol clarification.

Protocol clarification.


BOS161721 Boston Pharmaceuticals, Inc.


#### Section Description of Changes

#### Rationale

No longer

MAD data

collected has

been sufficient.

necessary for POC patients.

Section 6.2.1,

Laboratory Assessments, Table 2, Immunogenicity, PD and other Biomarker Tests column Add:

Immunogenicity, PD, and other Biomarker Tests

ADA nAb<sup>g</sup> pSTAT3 (predose Total IgG & IgM

Plasma CC Plasma CC

safety concerns.

pSTAT3 (predose [trough] samples only in Phase 1b)

& CCI

Whole blood for leukocyte immunophenotype (for MAD patients

only)
CCI
CCI
CRP

Direct Coomb's testh

Section 6.2.1.1, Pregnancy testing Replace:

Protocol clarification.

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, at the last follow up visit day (Day 270) and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures (see Section 5.4) are specified in the Schedule of Assessments (see Section 3.4).

With:

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, at the last follow up visit day (Day 270) and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures (see


BOS161721 Boston Pharmaceuticals, Inc.


#### Section Description of Changes

Rationale

Section 5.4) are specified in the Schedule of Assessments (see **Table 1** and **Table 4**).

Section 6.2.2.4, Causality of Adverse Events, Paragraph 1 Replace:

Protocol clarification.

The principal investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (**Table 4**) should be selected based on medical judgment, considering the definitions below and all contributing factors.

With:

The principal investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (**Table 3**) should be selected based on medical judgment, considering the definitions below and all contributing factors.

Section 6.2.3, Vital Signs

Replace:

Protocol clarification

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (Section 3.4). Vital signs will be assessed on Day 0 at predose and at Day 0, 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq 5$  minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

With:

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (**Table 1 and Table 4**). Vital signs will be assessed on Day 0 at predose and at Day 0, 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq 5$  minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

Section 6.2.4, 12-Lead Electrocardiogram, Paragraph 1

Replace:

Protocol clarification.

ECG will be assessed as specified in the Schedule of Assessments (Section 3.4). ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

With:

ECG will be assessed as specified in the Schedule of Assessments


BOS161721 Boston Pharmaceuticals, Inc.


#### Section **Description of Changes**

Rationale

(Table 1 and Table 4). ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

# Section 6.2.5,

Replace:

Protocol clarification.

Physical Examination, Paragraph 2

The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Section 3.4). It includes evaluation of patient complaints and SLE disease-related issues, and will exclude the genitourinary system.

With:

The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Table 1 and **Table 4**). It includes evaluation of patient complaints and SLE diseaserelated issues, and will exclude the genitourinary system.

#### Section 6.2.6,

C-SSRS, Paragraph 2

Replace:

Protocol clarification.

The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Section 3.4). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

With:

The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Table 1 and Table 4). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

#### Section 6.2.7, Injection Site Reactions

Replace:

Protocol clarification.

Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (Section 3.4). Local injection site reactions will be assessed at 2 hours postdose at baseline, and predose for each injection after baseline. Injection site reactions should be managed according to the standard of care. Injection site reactions, Grades 2 to 5, are to be reported as AEs of special interest (see Section 6.2.2.7.3).


#### Section Description of Changes

Rationale

With:

Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (**Table 1 and Table 4**). Local injection site reactions will be assessed at 2 hours postdose at baseline, and predose for each injection after baseline. Injection site reactions should be managed according to the standard of care. Injection site reactions, Grades 2 to 5, are to be reported as AEs of special interest (see Section 6.2.2.7.3).

Section 6.2.8, Immunogenicity, Paragraph 1 Replace:

Protocol clarification.

The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (Section 3.4). Blood samples (4 mL) to provide approximately 1.5 mL of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K2EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only analyzed by a central lab if the patient had a positive ADA on Day 90.

With:

The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (**Table 1 and Table 4**). Blood samples (4 mL) to provide approximately 1.5 mL of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K2EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only analyzed by a central lab if the patient had a positive ADA on Day 90.

Section 6.3, Efficacy Assessments Replace:

Protocol clarification.

All efficacy assessments will be performed at times defined in the Schedule of Assessments (Section 3.4).

With:

All efficacy assessments will be performed at times defined in the Schedule of Assessments (**Table 1 and Table 4**).

Section 6.4.2, PROs, Paragraph 1

Replace:

Protocol clarification.

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the CCI and the


#### Section

#### **Description of Changes**

Rationale

and will be assessed as specified in the Schedule of Assessments (Section 3.4).

With:

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the clinic and the and will be assessed as specified in the Schedule of Assessments (Table 1 and Table 4).

#### Section 6.5, Pharmacokinetic Assessments,

Paragraph 1

Replace:

Protocol clarification.

During the MAD Phase 1b (all sites) and POC Phase 2 (select sites only) parts of the study, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to Table 1 and Table 2.

With:

During the MAD Phase 1b (all sites) and POC Phase 2 (select sites only) parts of the study, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to **Table 4** and **Table 1**.

#### Section 6.6,

Pharmacodynamic Assessments, Paragraph 1 Replace:

Protocol clarification.

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (Section 3.4) for each of the following parameters:

With:

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (**Table 1 and Table 4**) for each of the following parameters:

### Section 6.6,

Pharmacodynamic Assessments, Bullet 5

#### Add:

Whole blood for leukocyte immunophenotype (for MAD patients only)

#### Section 7.4,

Accountability, Paragraph 1

#### Replace:

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Products returned to the pharmacy will be stored under the same conditions as products not yet dispensed.

No longer necessary for POC patients. MAD data collected has been sufficient. Clarification regarding handling of returned product.


BOS161721 Boston Pharmaceuticals, Inc.


#### Section

#### **Description of Changes**

Rationale

The returned products should be marked as 'returned' and kept separate from the products not yet dispensed.

With:

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Used investigational product returned to the pharmacy may be maintained in an ambient condition. Unused product should follow the instructions in the Pharmacy Manual. The used product that is returned should be marked as 'returned' and kept separate from the products not yet dispensed.

Section 8.2.1, Analysis Populations, Paragraph 1 Replace:

The primary efficacy analysis will be based on the FAS, defined as all patients who receive at least 1 dose of study treatment and at have least 1 evaluable post-baseline efficacy evaluation. FAS analyses will be conducted on the basis of the randomized treatment.

With:

The primary efficacy analysis will be based on the FAS, defined as all patients who receive at least 1 dose of study treatment and have **at** least 1 evaluable post-baseline efficacy evaluation. FAS analyses will be conducted on the basis of the randomized treatment.

Section 8.2.3, Primary Efficacy Endpoint(s), Paragraph 2

Add:

Patients that received prohibited medications or unallowable CS usage as described in Section 4.6 will be considered "medication failures" and will be treated as **statistical** non-responders **at the time points on or following the first date of prohibited medication or unallowable CS usage** for the primary efficacy analysis. The determination of medication failures will be reviewed using blinded data and finalized prior to unblinding.

Appendix 5 Replace:



Correction of typo.

Text added to address usage relative to analysis time points (ie patients are deemed nonresponders after usage but may still be responders prior to usage of prohibitive meds or CS). Clarification of active joint term.


Section Description of Changes Rationale




#### Section Description of Changes

Rationale



#### Appendix 7 Add:

Added for opioid dosing in SLE patients.

# ${\bf APPENDIX 9 \cdot OPIOID \cdot ORAL \cdot MORPHINE \cdot MILLIGRAM \cdot EQUIVALENTS \cdot OF \cdot COMMONLY \cdot USED \cdot OPIOIDS \P}$

| -Opioid·¤ | 30°mg·morphine·equivalent |
|--------------------------|---------------------------|
| -butorphanol¤ | 4.3·mg/day□ |
| -codeine¤ | 200·mg/day¤ |
| <u>dihydrocodeine</u> ¤ | 120·mg/dayo |
| •fentanyl·transdermal¤ | 12.5·mg/day¤ |
| •hydrocodone¤ | 30·mg/day□ |
| •hydromorphone¤ | 7.5·mg/day¤ |
| levorphanol tartrate¤ | 2.7·mg/day□ |
| meperidine· <u>HCl</u> ¤ | 300·mg/day¤ |
| oxycodone¤ | 20·mg/day¤ |
| <u>oxymorphone</u> ¤ | 10·mg/day¤ |
| -pentazocine¤ | 81.1·mg/day¤ |
| -tapentadol¤ | 75·mg/day¤ |
| tramadol¤ | 300·mg/day¤ |

Note that this list is not comprehensive. If an opioid is being used which is not in this list, please see the appropriate conversion factor below.


#### Section Description of Changes

Rationale

□ Opioid Oral Morphine Equivalent Conversion Factors a.b.

| Type of Opioid (strength in units) | MME Conversion Factor |
|---|---|
| Buprenorphine film/table <sup>c</sup> (mg) | 30 |
| Buprenorphine patch <sup>d</sup> (mcg/hr) | 12.6 |
| Buprenorphine film (mcg) | 0.03 |
| Butorphanol (mg) | 7 |
| Codeine (mg) | 0.15 |
| Dihydrocodeine (mg) | 0.25 |
| Fentanyl buccal or SL tablets, or lozenge/trochee (mcg) | 0.13 |
| Fentanyl film or oral spray <sup>f</sup> (mcg) | 0.18 |
| Fentanyl nasal spray <sup>g</sup> (mcg) | 0.16 |
| Fentanyl patch <sup>h</sup> (mcg) | 7.2 |
| Hydrocodone (mg) | 1 |
| Hydromorphone (mg) | 4 |
| Levorphanol tartrate (mg) | 11 |
| Meperidine hydrochloride (mg) | 0.1 |
| Methadone <sup>i</sup> (mg) | 3 |
| > 0, \le 20 | 4 |
| > 20, ≤ 40 | 8 |
| > 40, ≤ 60 | 10 |
| > 60 | 12 |
| Morphine (mg) | 1 |
| Opium (mg) | 1 |
| Oxycodone (mg) | 1.5 |
| Oxymorphone (mg) | 3 |
| Pentazocine (mg) | 0.37 |
| Tapentadol <sup>j</sup> (mg) | 0.4 |
| Tramadol (mg) | 0.1 |
| CDC = Centers for Disease Control: CMS = Centers for Medicare and | Medicaid Services: FDA = Food and |

CDC = Centers for Disease Control; CMS = Centers for Medicare and Medicaid Services; FDA = Food and Drug Administration; MAT = Medication Assisted Treatment; MME = morphine milligram equivalent; OMS = Overutilization Monitoring System.


BOS161721 Boston Pharmaceuticals, Inc.


#### **Description of Changes**

Rationale

- a. The MME conversion factor is intended only for analytic purposes where prescription data is used to calculate daily MME. It is to be used in the formula: Strength per Unit × (Number of Units/Days Supply) × MME conversion factor = MME/Day. This value does not constitute clinical guidance or recommendations for converting patients from one form of opioid analgesic to another. Please consult the manufacturer's full prescribing information for such guidance. Use of this file for the purposes of any clinical decision-making warrants caution.
- National Center for Injury Prevention and Control. CDC compilation of benzodiazepines, muscle relaxants, stimulants, zolpidem, and opioid analgesics with oral morphine milligram equivalent conversion factors, 2016 version. Atlanta, GA: Centers for Disease Control and Prevention; 2016. Available at https://www.cdc.gov/drugoverdose/media/. For more information, send an email to Mbohm@cdc.gov.
- Buprenorphine formulations with a FDA approved indication for MAT are excluded from Medicare's Overutilization Monitoring System's opioid overutilization reporting.

  The MME conversion factor for buprenorphine patches is based on the assumption that 1 milligram of
- The MME conversion factor for buprenorphine patches is based on the assumption that 1 milligram of parenteral buprenorphine is equivalent to 75 milligrams of oral morphine and that one patch delivers the dispensed micrograms per hour over a 24 hour day. Example:  $5 \mu g/hr$  buprenorphine patch × 24 hrs = 120 ug/day buprenorphine = 0.12 ug/day = 9 mg/day oral MME. In other words, the conversion factor not accounting for days of use would be 9/5 or 1.8. However, since the buprenorphine patch remains in place for 7 days, we have multiplied the conversion factor by 7 (1.8 × 7 = 12.6). In this example, MME/day for 4 5 µg/hr buprenorphine patches dispensed for use over 28 days would work out as follows: Example:  $5 \mu g/hr$  buprenorphine patch < (4 patches/28 days) × 12.6 = 9 MME/day. Please note that because this allowance has been made based on the typical dosage of 1 buprenorphine patch per 7 days, you should first change all Days Supply in your prescription data to follow this standard, i.e., Days Supply to buprenorphine patches x 7. data to follow this standard, i.e., Days Supply for buprenorphine patches = number of patches x ?
- The MME conversion factor for fentanyl buccal tablets, sublingual tablets, and lozenges/troche is 0.13. This conversion factor should be multiplied by the number of micrograms in a given tablet or lozenge/troche.
- lozenges/troche.

  The MME conversion factor for fentanyl film and oral spray is 0.18. This reflects a 40% greater bioavailability for films compared to lozenges/tablets and 38% greater bioavailability for oral sprays compared to lozenges/tablets.
- The MME conversion factor for fentanyl nasal spray is 0.16, which reflects a 20% greater bioavailability for sprays compared to lozenges/tablets.
- The MME conversion factor for fentanyl patches is based on the assumption that 1 milligram of parenteral fentanyl is equivalent to 100 milligrams of oral morphine and that 1 patch delivers the dispensed micrograms per hour over a 24 hour day. Example: 25  $\mu$ g/hr fentanyl patch × 24 hrs = 600 ug/day fentanyl = 60 mg/day oral morphine milligram equivalent.

  In other words, the conversion factor not accounting for days of use would be 60/25 or 2.4.

  However, since the fentanyl patch remains in place for 3 days, we have multiplied the conversion factor by 3 (2.4 × 3 = 7.2). In this example, MME/day for 10 25 µg/hr fentanyl patches dispensed for use over 30 days would work out as follows: Example:  $25 \mu g/hr$  fentanyl patch × (10 patches/30 days) × 7.2 = 60 MME/day. Please note that because
  - Example: 25 µg/hr fentanyl patch × (10 patches/30 days) × 7.2 = 60 MME/day. Please note that because this allowance has been made based on the typical dosage of 1 fentanyl patch per 3 days, you should first change all Days Supply in your prescription data to follow this standard, i.e., Days Supply for fentanyl patches = number of patches × 3.

    The CDC MME conversion factor to calculate morphine milligram equivalents is 3. CMS uses this conversion factor when analyzing Medicare population opioid use. CMS uses the graduated methadone MME conversion factors to calculate MME within the OMS for identifying and reporting potential opioid overutilizers. https://www.cdc.gov/drugoverdose/pdf/calculating\_total\_daily\_dose-a.pdf.

    Tapentadol is a mu receptor agonist and norepimephrine reuptake inhibitor. Oral MMEs are based on degree of mu-receptor agonist activity, but it is unknown if this drug is associated with overdose in the same dose-dependent manner as observed with medications that are solely mu receptor agonists.

same dose-dependent manner as observed with medications that are solely mu receptor agonists.

Add:

Appendix 8, Table 4

-Table 4 → Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| D | Screen*: | Enrolle | | | | Tre | eatment | Period: | Follow- | Upro | | | | Safet | y-Follow | -Upa |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28- | | 7-5 | 155 | 301 | 445 | 605 | 905 | 1205 | 1505 | 1805 | 1875 | 1955 | 2105 | 2405 | 2705 |
| Dayso | te~lo | 0a | (±%)c | (±13)o | (±%)0 | (±13)0 | (± <sup>1</sup> 3)0 | (±%)o | (±15)c | (±45)c | (± <sup>6</sup> 3)o | (±13)c | (±13)o | (±'5)o | (±13)o | (±°5): |
| Visit Numbero | lo | 2a | 0 | 3α | 40 | \$a | 6a | 70 | \$a | 9a | 10a | 0 | 0 | 11o | 12a | 13a |
| GENERAL-ASSESS | MENTS <sub>0</sub> | | | | | | | | | | | | | | | |
| Informed consents | Xo | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Inclusion/Exclusion<br>criteria: | Χo | п | 0 | | | | | | | | 0 | В | п | | | |
| • Medical history: | Χo | | 0 | п | | | 0 | | | | | 0 | 0 | | п | |
| Demographicso | Xo | | 0 | | | | 0 | | | | 0 | 0 | 0 | | | |
| SLICC Criteria for<br>SLE 10 | Xn | п | а | в | В | | | п | п | п | | а | а | | п | |
| Concomitant medication <sup>b</sup> o | Χo | Χn | Χo | Χo | Χn | Χo | Χα | Χn | Χn | Χn | Χo | Χo | Χn | Χn | Χn | Xo |
| Randomization's | | Xo | | | 0 | 0 | 0 | | | | 0 | | | 0 | | 0 |
| BOS161721 or<br>placebordosing u | | Xo | 0 | п | Xu | | Xo | Χn | Χn | Χo | Xu | 0 | 0 | | п | |
| SAFETY ASSESSM | ENTSo | | | | | | | | | | | | | | | |
| Full physical examo | Xo | Xo | 0 | в | 0 | 0 | 0 | а | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Chest'x-ray <sup>4</sup> 0 | Xo | 0 | 0 | | 0 | 0 | 0 | D | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| ·C-SSRSo | Xo | Xo | 0 | | | | 0 | Xn | | | Xo | 0 | 0 | | | |
| AEs and SAEso | | Xn | Xα | Xo | Xn | Xn | Xn | Χn | Χn | Χn | Xo | Xo | Xn | Xn | Xn | Χo |
| 12-lead ECG to | Xo | Xo | 0 | 0 | Xα | 0 | 0 | Χo | 0 | 0 | 0 | 0 | 0 | 0 | 0 | Xo |
| Injection site<br>reaction assessment | 0 | х6 | Xo | | Xo | | Xo | X <sub>0</sub> | Χo | Χo | Xo | Χo | Χo | Χo | Χo | Χo |
| Targeted physical examinations | 0 | а | п | Χo | Xo | Xo | Xo | X <sub>0</sub> | Χo | Χo | Xo | п | В | Χo | Χo | Χo |
| Vital signs (BP,<br>HR, and | | | а | | | | | | | | | О | О | | | |
| temperature) <sup>po</sup> | Xo | Xα | | Χn | Xα | Xα | Xα | Xo | Χo | Xα | Xα | | | Xn | Χn | Xo |
| · EFFICACY · ASSESS | | | | | | | | | | | | | | | | |
| BILAG-2004 Indexo | Xo | Xo | 0 | В | Xo | 0 | Xα | Xo | Xα | Χo | Xa | 0 | 0 | Xo | Xo | Xo |
| SLEDAI-2Klin | Xo | Χo | 0 | 0 | Χo | 0 | Xa | Xo | Χo | Χo | Xa | | | Χo | Χo | Χo |

Since Phase 1b MAD has completed, the Schedule of Assessments for Phase 1b MAD was moved to the Appendix.


#### Section Description of Changes

Rationale

| 0 | Screen*o | Enrollo | | | | Tre | atment | Period: | Follow- | Upm | | | | Safet | y Follow | -Upo |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7-5 | 159 | 30¶ | 445 | 60¶ | 90¶ | 1205 | 150¶ | 180¶ | 1875 | 1955 | 210¶ | 2405 | 270 |
| Dayso | to-la | 0a | (A <sup>4</sup> 1)c | (±3)0 | (#3)o | (±°3)a | (±°3)0 | (±°3)0 | (±'3)o | (±'5)0 | (±3)0 | (±3)a | (±°3)o | (±°3)a | (# <sup>3</sup> )o | (±'3): |
| Visit-Numbero | lo | 20 | 0 | 3a | 4a | 5a | 6a | 70 | 8a | 9a | 10a | 0 | 0 | 110 | 12a | 13a |
| ·PGA of disease | | | | | | | | | | | | 0 | | | | _ |
| activityo | Xα | Xo | | | Xο | | Xo | Xa | Xo | Χn | Xα | | | Xα | Xo | Xo |
| ACR-28-joint counts | Xα | Χn | 0 | В | Χn | | Xn | Xn | Xn | Χn | Χn | 0 | 0 | Χn | Xo | Xn |
| •CLASIo | Xo | Xo | | | Xo | | Xo | Xo | Xo | Xo | Χo | | 0 | Xo | Xo | Xo |
| CCI | 0 | Xα | 0 | В | Xo | 0 | Xo | Xo | Xo | Χo | Χo | 0 | 0 | Χo | Xo | Χo |
| ·SLICC/ACR· | | | 0 | | | | | | | | | 0 | 0 | | | _ |
| Damage Indexo | | Xα | | | | | | 0 | | | Χo | | | 0 | 0 | |
| CCI | | Χo | 0 | D | Xo | | Xo | Χn | Χo | Χn | Χn | 0 | 0 | Xα | Xo | Χn |
| LABORATORY ASS | ESSMEN | TSu | | | | | | | | | | | | | | |
| •CD4+-counts | Xα | Xα | 0 | Xo | Χo | Χo | а | Χa | в | 0 | Χo | 0 | 0 | в | 0 | 0 |
| ·Clinical laboratory | | | 0 | | | | | | | | | 0 | 0 | | | _ |
| assessments: | | | | | | | | | | | | | | | | |
| (hematology and | | | | | | | | | | | | | | | | |
| clinical chemistry)/o | Χū | Χn | | 0 | Χo | Χα | Χo | Xα | Xo | Xo | Χo | | | Xα | Xo | Xα |
| ·Coomb's test | | | 0 | | | | | | | | | 0 | 0 | | l l | |
| directio | Χn | Xo | | | Xo | | Χn | Χn | Xα | Χn | Xn<br>Xn | | $\longrightarrow$ | Xα | Xo | Χn |
| Total IgG and IgM to | Xo | Xo | 0 | Xo | Xo | Xo | 0 | Xo | 0 | 0 | 140 | 0 | 0 | 0 | 0 | 0 |
| Plasma CC | Χo | Χo | 0 | 0 | Χo | 0 | Χo | Xo | Xo | Χo | Χo | 0 | 0 | Χo | Xo | Χo |
| CCI | | | | | | | | | | | | 0 | | | | |
| | 0 | Xα | | Xο | Xα | 0 | Xα | Xα | 0 | 0 | Xα | | _ | 0 | 0 | 0 |
| Whole blood for | | | 0 | | | | | | | | | 0 | 0 | | | |
| leukocyte-<br>immunophenotypeo | | Χo | | Xo | Χo | | Χo | Χo | | | Χo | | | | | |
| ADA <sup>ke</sup> | 0 | Xn | | Xo | Xo | 0 | Xn | Xo | 0 | 0 | Xn | В | | 0 | 0 | Xn |
| nAbb | | 140 | | 160 | 140 | | 140 | Xo | - | - | Xo | 0 | | _ | _ | 140 |
| nSTAT3*0 | 0 | No. | | 0 | No. | No. | No. | Xo | | 0 | | _ | | 0 | 0 | 0 |
| | | Att | _ | D | All | Ao | Ass | .00 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| CCI | | Χo | 0 | Xo | в | | | Χo | | | Χn | 0 | 0 | | | Χo |
| | | | | | _ | _ | | | _ | _ | | _ | - | _ | _ | |
| | 0 | Χn | | D | | | п | В | D | 0 | 0 | D | | 0 | 0 | |

| 0 | Screen*o | Enrollo | | | | Tre | atment | Period: | Follow. | Up to | | | | Safet | y-Follow | -Upa |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dayso | -28-<br>to-lo | 0a | 74<br>(±91)o | 15¶<br>(±%)0 | 30¶<br>(±%)¤ | 44¶<br>(±%)o | 60¶<br>(±%)o | 90¶<br>(±%)o | 120¶<br>(±%)o | 150¶<br>(±%)o | 180¶<br>(±%)o | 187¶<br>(±%)0 | 195¶<br>(±%)o | 210¶<br>(±%)a | 240¶<br>(±%)o | 270¶<br>(±%): |
| Visit Numbero | lo | 20 | 0 | 30 | 40 | 5a | 6a | 7a | Sa . | 90 | 10a | 0 | 0 | 110 | 12a | 13a |
| CCI | | | п | | | | | | | | | п | D | | | |
| | Xo | Χu | | | Χo | | Xu | Χa | Χo | Xu | Xo | | | X*u | X*o | X*o |
| CRP0 | Xο | 0 | ū | 0 | D. | 0 | 0 | Xα | 0 | 0 | 0 | 10 | D | 0 | 0 | Xo |
| Serum pregnancy-<br>test (women): | Xn | | п | в | В | В | | В | В | в | ь | п | В | в | в | |
| FSH- | | | | | | | | | | | | | В | | | |
| (postmenopausal·<br>women):: | Xo | п | | | п | | | В | п | | | | | п | | |
| Urine pregnancy:<br>test (women)% | п | Χo | п | | Χo | | Xo | Χn | Χo | Χo | Χo | п | 0 | п | 0 | Χo |
| TB test<br>(QuantiFERON-<br>TB-Gold-In-Tube) <sup>4</sup> :: | Xo | а | ū | | D | 0 | 0 | 0 | D | | 0 | 0 | 0 | | а | |
| Serology (hepatitis:<br>Brand C, HIV-1/2:<br>combination) | Χo | | n | | | | | р | р | | | ū | В | | | |
| Stool nample <sup>p</sup> o | Xn | | | | | | - | | | | | | | | | - |
| Spot urine for protein/creatinine | | | п | | | | | | | | | 0 | D | | | |
| ration | Xo | Xσ | | 0 | Xn | р | Xa | Xσ | Xo | Xα | Xa | | | Xa | Xσ | Χo |
| Urinalysiso | Xn | Xn | 0 | | Xn | 0 | Xe | Xn | Xo | Xn | Xo | 0 | 0 | Xa | Xn | Xn |

| D | Screen*o | Enroll: Treatment Period Follow-Up to | | | | | | | | | | Safety Follow-Upo | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 74 | 155 | 305 | 445 | 605 | 905 | 1205 | 1505 | 180¶ | 1875 | 1955 | 210€ | 240¶ | 2705 |
| Dayso | to-la | 0 p | (49)0 | (±°3)o | (±93)a | (±°3)a | (49)0 | (±°3)0 | (#°3)a | (49)0 | (±°3)a | (±'3)a | (±°3)o | (#°3)0 | (±°3)0 | (4%)0 |
| Visit-Numbero | lo | 20 | 0 | 3a | 40 | 5a | 6a | 7a | 8a | 90 | 10a | D | O | llo | 12a | 13a |
| PK-Labso | | | | | | | | | | | | | _ | | | |
| Predosea | | Χα | 0 | | Xa | | Χα | Xo | Xo | Xa | Xo | | | 0 | D | п |
| Predose PK | | | D | | | | | | | | | 0 | 0 | | | |
| Windowa | 0 | 609ma | | 0 | ±:3%to | 0 | ±:39to | ±39da | ±3%0 | ±:3980 | ±3%0 | | | 0 | п | 0 |
| Postdosea | | X% | Χo | Xo | X40 | | | | | | X% | Χo | Χo | Xo | Xo | Xo |
| Postdose PK | | 4'h'±' | #"Ido | ±3°do | 4500 | | | | | | 4°h:±: | ±3*do | ±-3*do | ±3°da | ±3%0 | ±3'4: |
| Windowa | | 309m¶ | | | 30°m€ | | | | | | 30°m€ | | | | | |
| | | 8.p.+. | | | 83:4: | | | | | | 8°h±- | | | | | |
| | | 45°m¶ | | | 459m¶ | | | | | | 45°m¶ | | | | | |
| | | 24%·** | | | 24'h:+: | | | | | | 24h:±* | | | | | |
| | | 60°ma | | | 60°ma | | | | | | 60°mc | | | | | |
| immunodeficiency<br>neutralizing antib-<br>transcription 3; 5/<br>SLICC <sup>©</sup> Systemic<br>TDAR <sup>©</sup> T-cell dep | dy: PGA=T<br>AE=Serious:<br>Lupus Inter-<br>sendent antig | Physician<br>adverse e<br>national-<br>en respo | 's Glob<br>vent; S<br>Collabe<br>nse.¶ | al·Asses<br>C=Sub-<br>orating ( | sment; P<br>cutaneou<br>Clinics; | unoglobe<br>K pha<br>BC | din M: | IL-21= | interleu<br>STAT3 | kin 21;<br>≃°phos | IV=Int | ravenou<br>ed signa | s; m=1<br>l-transd<br><u>Act</u> ivity | rate; HI<br>ninute; n<br>ucer and<br>Index 20<br>tubercul | Ab=<br>activate<br>00; | |
| <ul> <li>Screening asset</li> <li>Concomitant v</li> <li>the daily dose</li> <li>further details</li> </ul> | ise of oral co<br>must be tape | rticostere | ids:∴A | maxim | ım-daily | dose of | | | | | | | | | | |
| <ul> <li>Grandomizatio</li> <li>Grandomizatio</li> <li>Fratients have screening. The months prior</li> <li>ECGs will be scheduled PK</li> </ul> | n should occu<br>e had a TB to<br>e vesults of T<br>o screening o<br>performed at | est and cl<br>B screen<br>or during<br>ter the pa | hest x r<br>ing, wh<br>the ser | ay withi<br>ich inclu<br>eening y | n 3 mont<br>des the t<br>period m | ths prior<br>QuantiF<br>ust be d | to scree<br>ERON®<br>scument | ning, th<br>TB-Gol<br>ed in st | en these<br>d In Tu<br>udy reco | rassessi<br>be (QF)<br>ords pri | nents do<br>F-G) test<br>or to ran | t and a c<br>adomiza | hest x-r<br>tion (Da | ay, cond<br>y 0).¶ | ncted in | the-3 |
| f - Injection sites | eaction asses | sments t | o be per | formed | at 2 hou | rs postd | 7.920 | | | | | | | | | |

•Table 4 - Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| D | Screen*0 | Enroll | hi Treatment Period Follow-Up to | | | | | | | | Safety-Follow-Up: | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 74 | 155 | 305 | 445 | 605 | 90€ | 1205 | 1505 | 180€ | 1875 | 195€ | 210€ | 2405 | 2705 |
| Dayso | to~lo | 0a | (tf1)o | (±15)a | (±93)a | (±°3)a | (±93)a | (±15)c | (±°3)0 | (±°3)a | (±°3)0 | (±°3)0 | (±°3)0 | (±°3)a | (±°3)0 | (±93)o |
| Visit:Numbero | 1o | 20 | 8 | 3α | 40 | 5a | 6a | 70 | 80 | 9a | 10a | 0 | 0 | 110 | 120 | 13a |
| 2 hours postdos | | | | | | | | | | | | | | | | |
| When the timin | g of these n | neasurem | emts coi | incides | rith a bl | ood-colle | ction, vi | ital sign | s should | be obta | ined pri | iortoth | etimerof | the bloc | od collec | tion. |
| h - SLEDAI-2K-the | ould-be-don | e-before: | random | ization | and dosi | ng-on-Da | sy@asrS | LEDAI | 2K < 6 | is exclu | sionary. | • | | | | |
| i → Clinical laborat | | | | | | | | | | | | | rhich wi | II-be mon | facting | • |
| → When clinically | | | | | | | | | | | | , | | | | |
| k - Blood samples only assayed (as | | | | | | | | ents."Su | bseque | nt ADA | samples | willber | collected | from al | l patient | s,·but· |
| 1 - nAbris collected | for all pati | ents, tho | ugh will | only-be | ranalyze | d by cen | traldab | if paties | atris pos | itive for | 'ADA'at | Day 90. | 4 | | | |
| =→ Predose (trough | ) samples | nly.¶ | _ | | | | | - | - | | | | | | | |
| a → Antibodies and | autoantibo | dies CC | | | | ill not be | e analyz | ed duri | ngsafet | y follow | upwisit | 1.4 | | | | |
| * - Urine pregnanc | | | | OCBP <sub>1</sub> | prior to: | tudy dry | ngradmi | nistrati | bravao | sing vis | its.¶ | | | | | |
| | | | | | | | | | | . " | - " | | | | | |


BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02




# A RANDOMIZED DOUBLE-BLIND PHASE 1b/2 COMBINED STAGGERED MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF LIMITED STANDARD OF CARE

**SPONSOR** Boston Pharmaceuticals, Inc.

55 Cambridge Parkway, Suite 400

Cambridge, MA 02142

United States of America (USA)

INVESTIGATIONAL COMPOUND: BOS161721

PROTOCOL NUMBER: BOS161721-02

PHASE Phase 1b/2

INVESTIGATIONAL NEW DRUG (IND) 131796

**NUMBER:** 


**VERSION NUMBER:** V5.0 (Amendment 4)

VERSION DATE: 23 January 2019


#### CLINICAL PROTOCOL APPROVAL FORM

| Protocol Title: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care | |
|---|---|
| Study Number: BOS161721-02 | |
| Version | Date |
| Original Protocol | 06 October 2017 |
| Protocol Version 2.0 (Amendment 1) | 14 November 2017 |
| Protocol Version 3.0 (Amendment 2) | 21 March 2018 |
| Protocol Version 4.0 (Amendment 3) | 27 July 2018 |
| Protocol Version 5.0 (Amendment 4) | 23 January 2019 |

This study protocol was subject to critical review and has been approved by sponsor. The information contained in this protocol is consistent with:

- The current risk-benefit evaluation of the investigational product.
- The moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (APPENDIX 2), and principles of Good Clinical Practices (GCP) as described in 21 Code of Federal Regulations (CFR) parts 50, 54, 56 and 312 and according to applicable local requirements.

The investigator will be supplied with details of any significant or new findings, including adverse events, relating to treatment with the investigational product.

I agree with these statements and indicate my approval by signature for this protocol:

| Name and Title | Signature and Date |
|---|---|
| PPD MD, PhD Chief Medical Officer Boston Pharmaceuticals | PPD |
| PPD MD, FACR Vice President, Clinical Development Boston Pharmaceuticals | PPD |
| PPD Clinical Operations Lead Boston Pharmaceuticals | PPD ' |
| PPD MD, PhD Vice President, Clinical Development and Safety Officer Boston Pharmaceuticals | PPD |


#### BOS161721-02

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

#### CONFIDENTIALITY AND INVESTIGATOR STATEMENT

The information contained in this protocol and all other information relevant to BOS161721 are the confidential and proprietary information of Boston Pharmaceuticals, Inc., and except as may be required by federal, state, or local laws or regulation, may not be disclosed to others without prior written permission of Boston Pharmaceuticals, Inc.

I have read the protocol (Version 5.0, dated 23 January 2019), including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described. I will conduct this study as outlined herein, in accordance with the regulations stated in the Federal Code of Regulations for Good Clinical Practices and International Council for Harmonisation (ICH) guidelines, and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and any amendments, and access to all information provided by Boston Pharmaceuticals, Inc., or specified designees. I will discuss the material with them to ensure that they are fully informed about BOS161721 and the study.

| Principal In | nvestigator Name (printed) | Signature |
|--------------|----------------------------|-----------|
| Date | Site Number | |


# PROTOCOL SUMMARY

| Title: | A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care |
|---|---|
| Indication | Adults with moderately to severely active SLE |
| Background and Rationale | SLE is a chronic systemic autoimmune disease with considerable heterogeneity in clinical manifestations and disease course. There is evidence that B- and T-cells are critical to the development of the disease, and that T-cell-derived cytokines such as interleukin-21 (IL-21) are involved in the SLE-associated inflammatory pathological response. |
| | BOS161721 is a humanized immunoglobulin G1 (IgG1) triple mutation monoclonal antibody (mAb) intended to have an extended terminal elimination half-life (t½) that selectively binds to and neutralizes IL-21, which acts on multiple cell types that drive inflammation and autoimmunity. <i>In vivo</i> , BOS161721 inhibits T-cell dependent antigen responses of B-cells and is being developed as a potential treatment for adults with moderately to severely active SLE. |
| | Nonclinical studies have evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), pharmacokinetics (PK), and immunogenicity of BOS161721 administered intravenously (IV) and subcutaneously (SC). The no observed adverse effect level (NOAEL) in Cynomolgus monkeys was determined to be 100 mg/kg (SC and IV), the highest dose tested. There were no injection site reactions in animals dosed subcutaneously. |
| | In a Phase 1 single ascending dose (SAD) study, BOS161721 was administered IV and SC to healthy male and female adult subjects. This double-blind, placebo-controlled study evaluated 8 ascending dose levels (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) for safety, tolerability, PK, PD and immunogenicity. Overall, there were no clinically significant safety or tolerability findings from this study. |
| | Results from the Phase 1 SAD study informed the dose regimens used for the multiple ascending doses (MAD) Phase 1b portion of this trial. The MAD portion will involve 3 cohorts. The Phase 2 portion will be a proof of concept (POC) part, where dose selection will be based on the data monitoring committee (DMC) and sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD portion of 30 patients treated with BOS161721/placebo. The purpose of the study is to establish a safe and effective dosage for adult patients with moderately to severely active SLE. |


BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02


# **Objectives and Endpoints:**

#### **MAD Phase 1b**

Primary

## Safety Endpoints

relatedness

# • To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose.

**OBJECTIVES** 

 Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and

**ENDPOINTS** 

- Injection site reactions
- Columbia Suicide Severity Rating Scale (C-SSRS)
- 12-lead electrocardiograms (ECGs) parameter results at each visit and change from baseline
- Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline
- Clinical laboratory results and change from baseline
- Physical examinations changes from baseline
- Anti-drug antibodies (ADAs)
- Study drug exposure/compliance

#### **Secondary**

 To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PD effects in patients with moderately to severely active SLE.

#### Pharmacokinetic Endpoints

- BOS161721 concentration by visit and time point
- Maximum observed concentration (C<sub>max</sub>), first time to maximum concentration (T<sub>max</sub>), area under the concentration-time curve (AUC), t<sub>1/2</sub>, systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>)

#### Pharmacodynamic Endpoints

- Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype
- Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit
- Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit





BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02


#### **POC Phase 2**

#### **OBJECTIVES ENDPOINTS Primary** Primary Efficacy Endpoint To demonstrate a superior effect of BOS161721 at the chosen dose The proportion of patients with a SRI-4 response at Day 210 (see Section 6.3.4.1) compared with placebo for response on the SLE Responder Index 4 (SRI-4) Secondary Secondary Efficacy Endpoints To demonstrate a superior effect of BOS161721 at the chosen dose The proportion of patients with: compared with placebo for SRI-4 response at each visit response on clinical indicators of SRI-5 and SRI-6 response at each visit SLE activity, in adult patients with (Section 6.3.4.2) moderately to severely active SLE a sustained reduction of oral on limited background standard of corticosteroid (CS) (< 10 mg/day and care treatment ≤ Day 0 dose) between Day 120 and Day 210 new BILAG A flare or > 1 BILAG B flares relative to baseline through Day 210 PGA worsening a BICLA response a CLASI response medication failures Results and changes from baseline in: **CLASI** swollen and tender joints ACR-28 SLEDAI-2K SLICC/ACR damage index Time to medication failure Duration of longest SRI-4 response Time to first SRI-4 response Time to BILAG A flare or > 1 BILAG B flare compared to baseline through Day 210 **Safety** To assess safety and tolerability of Safety Endpoints repeat doses of BOS161721 at the Incidence and severity of adverse events chosen dose administered SC in (AEs) and serious adverse events (SAEs), adult patients with moderately to related AEs, AEs leading to study drug severely active SLE on limited discontinuation, AEs by severity and background standard of care relatedness treatment Injection site reactions C-SSRS 12-lead ECGs parameter results at each visit and change from baseline Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline Clinical laboratory results and change from




#### **Study Design:**

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of multiple SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, eligible patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly. The trial will consist of 2 double-blinded portions: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

The MAD Phase 1b portion of the study design will consist of 3 cohorts, with Cohort 1 containing 6 patients, where 5 of these patients will receive BOS161721 (active), and 1 will receive placebo. Cohorts 2 and 3 will each contain 12 patients, including 9 active and 3 placebo patients. Dose selection for each cohort is based on 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. Each of the 3 doses (20, 60, and 120 mg) selected for the MAD portion are projected not to exceed the mean exposure of that achieved in the SAD study following the single 240 mg SC dose. Each patient may receive a total of


7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

The MAD portion design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after the DMC evaluates the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after the DMC evaluation of the safety and tolerability data from Cohort 2 and Cohort 1. Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. This dose will not exceed doses tested during the MAD portion.

For the POC portion, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio. As in the MAD portion, each patient in the POC portion may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 60. Tapering of steroids during the course of the study will be highly encouraged and should be evaluated at the protocol permitted visits (Day 0 through Day 60 and Day 120 through Day 150). Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant due to the endpoint evaluations occurring at Day 120 and Day 210.

DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.


#### Main Criteria for Inclusion and Exclusion

#### **Inclusion Criteria:**

1. Men and women, ages 18 to 70 years, inclusive

- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion OR Lupus nephritis as the sole clinical criterion in the presence of antinuclear antibodies [ANA] or anti- double-stranded deoxyribonucleic acid [dsDNA] antibodies), either sequentially or simultaneously
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
  - c. C3 or C4 levels below normal as determined by the central lab
- 5. At screening, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA,


decreased complement, thrombocytopenia, and leukopenia

- ii. Points from lupus headache and organic brain syndrome will also be excluded
- 7. Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 4.4

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization)
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment


with study drug plus 52 weeks

11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

#### **Exclusion Criteria**

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic sclerosis, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed


8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study

- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count < 350/μL at screening
- 16. Platelets < 50,000/mm<sup>3</sup> (50  $\times$  10<sup>9</sup>/L) or < 35,000/ mm<sup>3</sup> (35  $\times$  10<sup>9</sup>/L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation
- 20. Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) > 2 × the upper limit of normal (ULN) at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK) > 3.0 × ULN at screening unless related to lupus myositis
- 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic mAb (eg, IgG protein) or molecules made of components of mAbs
- 25. History substance and/or alcohol abuse, or dependence within the past 1


year, at the investigator's judgment

26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision)

- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 on the C-SSRS
- 31. Current or pending incarceration
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness

## Statistical Considerations

Below is a summary of the statistical methods. Further details can be found in Section 8.

Two analyses are planned: 1) an interim analysis to select the POC dose based on the MAD data, and 2) a final analysis at study completion. Additionally, DMC safety analyses will be performed for each MAD cohort and throughout the POC to monitor patient safety as described in the DMC charter. An additional analysis may be performed for the MAD portion of the study when all MAD patients have completed the safety follow-up, or withdrawn from the study, and prior to the final analysis. Data from the POC part of the study will be excluded from this additional analysis.

Unless stated otherwise, statistical testing will only be performed on the POC data and will be done using 2-sided overall alpha of 0.10. Data will be summarized descriptively by treatment and overall for each study phase. For the MAD portion, BOS161721 will be summarized overall and by each dose level and placebo patients from each cohort will be combined.

The descriptive summaries for the categorical data will include number and percentage. The descriptive summaries for the continuous data will include number, mean, median, standard deviations (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles,


minimum, median, and maximum. Counts, medians, 25<sup>th</sup> and 75<sup>th</sup> percentiles, and standard error will be presented for time-to-event data.

All safety analyses will be performed using the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. All efficacy analyses will be performed using the full analysis set (FAS), defined as all patients who receive at least 1 dose of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. Select efficacy analyses may also be performed on the per protocol (PP) set.

Binary efficacy endpoints, including the primary efficacy endpoint, will be assessed via Pearson's chi-squared analysis.

Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) when applicable, adjusting for the baseline value. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test.

Adverse event data will be coded to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be summarized, based on coded terms, using frequency and percentage of patients. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters, will be summarized at each individual visit.


Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 23 January 2019; V5.0

# **TABLE OF CONTENTS**

| CLINICAL PROTOCOL APPROVAL FORM | 2 |
|--------------------------------------------------------|----|
| CONFIDENTIALITY AND INVESTIGATOR STATEMENT | 3 |
| PROTOCOL SUMMARY | 4 |
| TABLE OF CONTENTS | 16 |
| LIST OF IN-TEXT TABLES | 19 |
| LIST OF IN-TEXT FIGURES | 19 |
| LIST OF ABBREVIATIONS | 20 |
| 1. INTRODUCTION AND RATIONALE | 24 |
| 1.1 Indication | |
| 1.2 Background and Rationale | 24 |
| 1.2.1 Overview of the Disease State | 24 |
| 1.2.2 BOS161721 Development | 24 |
| 1.2.2.1 Interleukin-21 | 25 |
| 1.2.2.2 Preclinical Studies | |
| 1.2.2.3 Clinical Studies | |
| 1.2.3 Study Dose Selection | 28 |
| 1.2.4 Risk-Benefit Assessment | 29 |
| 1.2.5 Potential Risks | |
| 1.2.5.1 Anaphylaxis and Serious Allergic Reactions | |
| 1.2.5.2 Injection Site Reactions | 31 |
| 1.2.5.3 Immune Complex Disease | |
| 1.2.5.4 Infections | |
| 1.2.5.5 Malignancy | 33 |
| 1.2.5.6 Hepatic Function Abnormality | |
| 1.2.5.7 Failure of Vaccination | |
| 1.2.5.8 Potential for Drug-Drug Interactions | |
| 1.2.5.9 Potential Risk to Fetal Development | |
| 2 STUDY OBJECTIVES AND ENDPOINTS | |
| 2.1 Phase 1b Multiple Ascending Dose | |
| 2.2 Phase 2 Proof of Concept | |
| 3 STUDY PLAN | |
| 3.1 Study Design | |
| 3.1.1 Multiple Ascending Dose Phase 1b | |
| 3.1.1.1 Dose Escalation for the MAD Portion | |
| 3.1.1.2 Dose Limiting Toxicity (DLT) | |
| 3.1.1.3 DMC Recommendations | |
| 3.1.2 POC Phase 2 | |
| 3.1.2.1 BOS161721 POC Dose Selection and Justification | 39 |

| Clinical | Study | Protocol: | DOC1 | 61721 | $\Omega$ |
|----------|-------|-----------|------|-------|----------|
| Ciinicai | Stuav | Protocor: | BOST | 01/21 | -02 |

| Protocol Date an | d Version: 23 | 3 January | z 2019: V5.0 |
|------------------|---------------|-----------|--------------|
|------------------|---------------|-----------|--------------|

| 3.1.2. | POC Study Design | 40 |
|--------|-------------------------------------------------------------|----|
| 3.2 | Randomization and Blinding | 40 |
| 3.3 | Study Schematic | 42 |
| 3.4 | Schedule of Assessments | 43 |
| 3.5 | End of Study | 52 |
| 4 P | OPULATION | 52 |
| 4.1 | Participant Recruitment | 52 |
| 4.2 | Number of Patients | 52 |
| 4.3 | Patient Screening | 52 |
| 4.4 | Inclusion Criteria | 52 |
| 4.5 | Exclusion Criteria | 54 |
| 4.6 | Concomitant Medications | 57 |
| 4.6.1 | Corticosteroid | 57 |
| 4.6.2 | Other Prohibited and/or Restricted Treatments | 58 |
| 4.7 | Women of Childbearing Potential | 58 |
| 4.7.1 | Determination of Menopause | 59 |
| 4.7.2 | Contraception | 59 |
| 4.8 | Deviation from Inclusion/Exclusion Criteria | 59 |
| 4.8.1 | Patient Withdrawal and Replacement | 60 |
| 5 S | TUDY PROCEDURES | 60 |
| 5.1 | Screening | 60 |
| 5.1.1 | Retesting During Screening Period | 61 |
| 5.2 | Enrollment/Randomization and Day 0 Treatment | 61 |
| 5.3 | Treatment Period/Follow-Up Visits | 62 |
| 5.4 | Safety Follow-Up Visits | 63 |
| 5.5 | Premature Discontinuation. | 64 |
| 6 A | ASSESSMENTS | 64 |
| 6.1 | Medical History, Demographic and Other Baseline Information | 65 |
| 6.2 | Safety Assessments | 65 |
| 6.2.1 | Laboratory Assessments | 65 |
| 6.2.1. | 1 Pregnancy testing | 67 |
| 6.2.1. | 2 Tuberculosis Screening | 67 |
| 6.2.2 | Adverse Events | 68 |
| 6.2.2. | 1 Definitions | 68 |
| 6.2.2. | 2 Recording of Adverse Events | 68 |
| 6.2.2. | 3 Severity of Adverse Events | 68 |
| 6.2.2. | 4 Causality of Adverse Events | 68 |
| 6.2.2. | 5 Seriousness of Adverse Events | 69 |
| 6.2.2. | 6 Adverse Events of Special Interest | 70 |
| 6.2.2. | 7 Reporting of Adverse Events | 73 |
| 6.2.2. | 8 Follow Up of Adverse Events | 75 |

| Clinical | Study | Protocol: | DOC1 | 61721 | $\Omega$ |
|----------|-------|-----------|------|-------|----------|
| Ciinicai | Stuav | Protocor: | BOST | 01/21 | -02 |

| FIOLOCO | Date and Version. 25 January 2019, V5.0 | |
|---------|--------------------------------------------------------------|----|
| 6.2.3 | Vital Signs | 75 |
| 6.2.4 | 12-Lead Electrocardiograms | |
| 6.2.5 | Physical Examinations | 76 |
| 6.2.6 | C-SSRS | 76 |
| 6.2.7 | Injection Site Reactions | 76 |
| 6.2.8 | Immunogenicity | 76 |
| 6.3 | Efficacy Assessments | 77 |
| 6.3.1 | SLEDAI-2K | 77 |
| 6.3.2 | BILAG 2004 | 77 |
| 6.3.3 | PGA of Disease Activity | 77 |
| 6.3.4 | Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response | 78 |
| 6.3.4.1 | | |
| 6.3.4.2 | SRI-5 and SRI-6 Response | 78 |
| 6.3.4.3 | BICLA Response | 78 |
| 6.3.5 | CLASI Response | 78 |
| 6.3.6 | ACR-28 Joint Count | 79 |
| 6.4 | Other Variables | 79 |
| 6.4.1 | SLICC/ACR Damage Index | 79 |
| 6.4.2 | PROs | 79 |
| 6.5 | Pharmacokinetic Assessments | 79 |
| 6.6 | Pharmacodynamic Assessments | 79 |
| 6.7 | Pharmacokinetic/Pharmacodynamic Relationship | 80 |
| 6.8 | Protocol Deviations | 80 |
| 7 S | ΓUDY DRUG MANAGEMENT | 80 |
| 7.1 | Description | 80 |
| 7.1.1 | Formulation | 80 |
| 7.1.2 | Storage | 80 |
| 7.2 | Packaging and Shipment | 80 |
| 7.3 | Dose and Administration | 80 |
| 7.4 | Accountability | 81 |
| 7.5 | Prohibited Concomitant Therapy | 81 |
| 7.6 | Compliance | 81 |
| 8 S | TATISTICS | 81 |
| 8.1 | Sample Size | 82 |
| 8.2 | Statistical Methods | 83 |
| 8.2.1 | Analysis Populations | 83 |
| 8.2.2 | Demographics and Baseline Characteristics | 83 |
| 8.2.3 | Primary Efficacy Endpoint(s) | 83 |
| 8.2.4 | Secondary Efficacy Endpoint(s) | 84 |
| 8.2.5 | Analysis of Safety | 84 |
| 8.2.5.1 | Safety Analysis | 84 |

| Clinical Study Protocol: | ROS161721-02 |
|--------------------------|--------------|

| 8.2.6 Ph | armacokinetic and Pharmacodynamic Data | 84 |
|---|---|---|
| 8.2.6.1 | Analysis of Pharmacokinetic Data | 84 |
| 8.2.6.2 | Analysis of Pharmacodynamic Data | 85 |
| 8.2.6.3 | Population Pharmacokinetic Analysis or PK/PD Modeling | 85 |
| 8.3 Interir | n Analysis and Power | 85 |
| 9 ETHICS | AND RESPONSIBILITIES | 85 |
| 9.1 Good | Clinical Practice | 85 |
| 9.2 DMC | | 85 |
| 9.3 Institu | tional Review Board/Independent Ethics Committee | 86 |
| 9.4 Inform | ned Consent | 86 |
| 9.5 Recor | ds Management | 87 |
| 9.6 Source | e Documentation | 88 |
| 9.7 Study | Files and Record Retention. | 88 |
| 10 AUDITI | NG AND MONITORING | 88 |
| 11 AMEND | MENTS | 88 |
| 12 STUDY | REPORT AND PUBLICATIONS | 89 |
| 13 STUDY | DISCONTINUATION | 89 |
| 14 CONFID | ENTIALITY | 89 |
| 15 REFERE | NCES | 91 |
| 16 APPEND | DICES | |
| APPENDIX 1 | NAMES OF STUDY PERSONNEL | 95 |
| APPENDIX 2 | DECLARATION OF HELSINKI | 96 |
| APPENDIX 3 | | |
| APPENDIX 4 | MEDICATION WASHOUT PERIODS | 101 |
| APPENDIX 5 | BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA) | 102 |
| APPENDIX 6 | INJECTION SITE REACTION GRADING SCALE | 103 |
| APPENDIX 7 | PROTOCOL SUMMARY OF CHANGES | 104 |
| | LIST OF IN-TEXT TABLES | |
| Table 1. | Schedule of Assessments - Phase 1b - Multiple Ascending Dose | 43 |
| Table 2. | Schedule of Assessments - Phase 2 Proof of Concept (POC) | |
| Table 3. | Laboratory Tests | |
| Table 4. | Causality Definitions | |
| | LIST OF IN-TEXT FIGURES | |
| Figure 1. | Individual pSTAT3 C <sub>min</sub> Levels Versus Dose | 29 |
| Figure 2. | Study Diagram for MAD Phase 1b and POC Phase 2 | |


## LIST OF ABBREVIATIONS

ACR American College of Rheumatology

ADA anti-drug antibody
AE adverse event

AIDS acquired immune deficiency syndrome

ALT alanine aminotransferase
ANA antinuclear antibodies
ANC absolute neutrophil count
ANOVA analysis of variance
ANCOVA analysis of covariance
APL antiphospholipid

AST aspartate aminotransferase

AUC area under the concentration-time curve

AZA azathioprine

BICLA BILAG-based Composite Lupus Assessment

BILAG British Isles Lupus Assessment Group

BP blood pressure BUN blood urea nitrogen

BW body weight C complement

C-SSRS Columbia Suicide Severity Rating Scale

CD cluster of differentiation

CK creatine kinase
CL systematic clearance

CLASI Cutaneous Lupus Erythematosus Area and Severity Index

C<sub>max</sub> maximum plasma concentration

CMH Cochran-Mantel-Haenszel

CS corticosteroids

CSR clinical study report
DILI drug-induced liver injury
DLT dose-limiting toxicity
DMC data monitoring committee

dsDNA double-stranded deoxyribonucleic acid

ECG electrocardiogram
EOT end of treatment

eCRF electronic case report form

F female

CCI

FAS full analysis set

Fc fragment crystallizable


Clinical Study Protocol: BOS161721-02


FDA Food and Drug Administration FSH follicle stimulating hormone GCP Good Clinical Practice

eGFR estimated glomerular filtration rate

GLP Good Laboratory Practice

GWAS genome-wide association studies

γc gamma chain HBV hepatitis B virus

hCG human chorionic gonadotropin

HCl hydrochloride HCV hepatitis C virus

HIV human immunodeficiency virus

HR heart rate

HRT hormone replacement therapy

IA interim analysis

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonization

IEC Independent Ethics Committee

Ig immunoglobulin
IL interleukin

IL-21R interleukin 21 receptor

IM intramuscular IFNγ interferon gamma

INR International Normalized Ratio
IRB Institutional Review Board

IUD intrauterine device

IV intravenous

IVRS interactive voice response system

JAK Janus kinase kg kilogram

KLH keyhole limpet hemocyanin LOCF last observation carried forward

M male

mAb monoclonal antibody
MAD multiple ascending dose

MAPK mitogen-activated protein kinase

MedDRA Medical Dictionary of Regulatory Activities

MS multiple sclerosis MTX methotrexate

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events


Clinical Study Protocol: BOS161721-02


NIAID/FAAN National Institute of Allergy and Infectious Diseases/Food Allergy and

Anaphylaxis Network

NK natural killer

NOAEL no observed adverse event level

NO nitric oxide

OTC over-the-counter
PD pharmacodynamics
PEF peak expiratory flow

PGA Physician's Global Assessment

PK pharmacokinetics
POC proof of concept
PP per protocol

PR (interval) from onset of the p-wave to the end of the r-wave

pSS primary Sjögren's syndrome

pSTAT3 phosphorylated signal transducer and activator of transcription 3

PT preferred term

QRS (interval) from the onset of the q-wave to the end of the s-wave
QT (interval) from onset of the QRS complex to the end of the T wave
QTcF QT interval corrected for heart rate using Fridericia's formula

QFT-G QuantiFERON-TB Gold In-Tube

RA rheumatoid arthritis

RR (interval) from the onset of the r-wave to the onset of the next consecutive r-

wave

SAD single ascending dose SAE serious adverse event SAP statistical analysis plan

SC subcutaneous

SDMT safety data monitoring board

CCI

SLE systemic lupus erythematosus SLEDAI-2K SLE Disease Activity Index 2000

SLICC Systemic Lupus International Collaborating Clinics

Sm Smith

SOC system organ class
SRI-4 SLE Responder Index 4
SRI-5 SLE Responder Index 5
SRI-6 SLE Responder Index 6
SS safety analysis set

SSA Sjögren syndrome-A (Ro) SSB Sjögren syndrome-B (La)

STAT3 signal transducer and activator of transcription 3


Clinical Study Protocol: BOS161721-02


SUSAR suspected unexpected serious adverse reaction

ty<sub>2</sub> terminal elimination half-life

TB tuberculosis

TDAR T-cell dependent antibody response

Tfh T-follicular helper

Th T-helper

TK toxicokinetics

T<sub>max</sub> first time to maximum concentration

Treg regulatory T-cell
ULN upper limit of normal

US United States

Vd volume of distribution

WBC white blood cell

WHO World Health Organization
WOCBP women of childbearing potential

YTE triple mutation


## 1. INTRODUCTION AND RATIONALE

#### 1.1 Indication

BOS161721 is a humanized monoclonal antibody (mAb), which binds to and inhibits interleukin-21 (IL-21) bioactivity, and is being developed for the treatment of moderately to severely active systemic lupus erythematosus (SLE) in adults.

## **1.2** Background and Rationale

#### 1.2.1 Overview of the Disease State

SLE is a chronic inflammatory autoimmune disease that has variable manifestations in multiple organ systems and follows a relapsing and remitting course. The disease process includes abnormal immune responses mediated by tissue-binding autoantibodies and immune complex deposition, giving rise to tissue damage often resulting in end organ disease and even mortality. Survival of SLE has improved due to earlier detection, improved overall medical care, and standardized SLE treatment with corticosteroids (CS), immunosuppressants, and cytotoxic agents. However, some of the morbidity in patients with SLE is related to its treatment. Comparison of early and late outcomes in patients with SLE demonstrate that death in early disease is most commonly due to infections and active SLE causing multi-system organ damage, while thromboses were the most common cause of death during later disease.<sup>2</sup>

The reported prevalence of SLE in the United States (US) is 20 to 70 cases per 100,000 people.<sup>3</sup> More than 90% of cases of SLE occur in women, frequently starting at childbearing age. Women of color are disproportionately affected by SLE. This suggests multiple genetic and environmental factors are at play. Accordingly, a multifactorial view of the immunopathogenesis of SLE suggests more than 1 area of interest, including breach in central tolerance in the adaptive arm of the immune system, peripheral amplification of the autoimmune response by the innate immune system, and local processes in the target organ that facilitate end-organ disease.<sup>4</sup>

#### **1.2.2 BOS161721 Development**

Boston Pharmaceuticals is developing BOS161721 for the treatment of SLE. BOS161721 is a humanized immunoglobulin G1 (IgG1) mAb with extended half-life directed against human IL-21.

Murine mAb 19E3, the progenitor of BOS161721, was generated using mouse hybridoma technology. 19E3 has subpicomolar (pM) affinity to human IL-21 and was selected for its potent neutralization of IL-21 bioactivity. BOS161721 was generated by the humanization of mAb 19E3 where its complementarity-determining regions were grafted onto a human IgG1 kappa backbone. The fragment crystallizable (Fc) portion of BOS161721 contains a YTE (M252Y/S254T/T256E triple mutation) in the constant domain of the IgG1 heavy chain that was introduced into the parental molecule, 19E3, intended to prolong the *in vivo* terminal elimination half-life (t½) of the mAb. Thus, BOS161721 retains sub-pM binding to IL-21 and prevents IL-21 from binding to the IL-21 receptor (IL-21R), inhibiting IL-21 bioactivity.


BOS161721 binds to human IL-21 and Cynomolgus monkey IL-21, which are highly homologous, and neutralizes the bioactivity of both. BOS161721 is specific for IL-21 as it does not bind to or inhibit the other gamma-chain (γc) family of cytokines, and acts to specifically neutralize the IL-21 pathway. In *in vitro* studies, BOS161721 inhibited downstream IL-21-induced signaling, IL-21-induced plasma cell differentiation, and IL-21-induced natural killer (NK) cell activation. In *in vivo* studies, BOS161721 significantly inhibited the T-cell dependent antibody response (TDAR) to immunization with a protein antigen as well as B-cell expansion following a second protein antigen immunization in Cynomolgus monkeys.

#### **1.2.2.1 Interleukin-21**

IL-21 is an inflammatory cytokine, which belongs to a family of cytokines that also includes IL-2, IL-4, IL-7, IL-9, and IL-15, all of which bind to private receptors in complex with the common cytokine receptor yc. 6 Most cytokines in this family are critically important for both the maintenance and function of T-cell and B-cell responses. IL-21 signals through a receptor complex consisting of its own private receptor, the IL-21R and vc.<sup>6,7</sup> Engagement of the IL-21R/γc complex leads to the activation of several signaling pathways, including the Janus kinase/signal transducer and activator of transcription, mitogen-activated protein kinase (MAPK) and phosphoinositide 3-kinase pathways. EL-21 is produced mainly by T-cells and NK T-cells, but neutrophils have also been reported to produce IL-21. 9,10 The IL-21R is expressed on a broad array of cell types, including B-cells, T-cells, NK-cells, macrophages and dendritic cells, as well as other hematopoietic and nonhematopoietic cells such as fibroblasts, keratinocytes, and intestinal epithelial cells.<sup>9,11</sup> Activation of signal transducer and activator of transcription 3 (STAT3) via phosphorylation is critical in regulating human B-cell responses to IL-21<sup>12</sup>; phosphorylated STAT3 (pSTAT3) forms a homodimer, which translocates to the nucleus where it initiates transcription of the IL-21 gene, forming an autocrine loop for IL-21 production via STAT3 phosphorylation. <sup>13</sup> In addition, IL-21 has been shown to upregulate expression of its own receptor <sup>14</sup> and induces an autocrine feedback loop. <sup>15</sup>

IL-21 modulates various aspects of immune function. It promotes cluster of differentiation 4 (CD4+) T-cell differentiation and promotes the generation of T-helper (Th)17<sup>16</sup> and T-follicular helper (Tfh) cells. <sup>15,17</sup> In mice, IL-21 has been shown to regulate the balance between Th17 and regulatory T-cell (Treg), in that it increases Th17, while inhibiting Treg differentiation. <sup>18</sup> Less is understood with regards to human Tregs, although IL-21 has been reported to counteract Treg suppression of human effector T-cells <sup>19</sup> and blockade of IL-21 promotes Treg generation in a murine model of graft versus host disease induced by human T-cells. <sup>20</sup> IL-21 upregulates CD8+ T-cell and NK-cell expansion and cytolytic activity by increasing granzyme B and perforin. <sup>21,22</sup> IL-21 also has been reported to increase granzyme B in plasmacytoid dendritic cells and B-cells resulting in inhibition of T-cell responses. <sup>23,24</sup> IL-21 also has a variety of effects on nonhematopoietic cells, such as stromal cells and induces inflammation through matrix metalloproteinase release by gut intestinal fibroblasts. <sup>25</sup>

One principal non-redundant role of IL-21 is the promotion of B-cell activation, differentiation, or death during humoral immune responses. <sup>14</sup> Furthermore, increased IL-21 production is characteristic of several autoimmune diseases and is likely to contribute to autoantibody production as well as pathologic features of autoimmune disease. <sup>26</sup> The critical role of IL-21 in promoting humoral and other immune responses makes it an important focus of potential


Clinical Study Protocol: BOS161721-02


therapeutic interventions in conditions characterized by overproduction of pathogenic autoantibodies. IL-21 production by Tfh cells in humans is believed to play a major role in driving the autoantibody production through its role in plasma cell differentiation. Importantly, Tfh cell populations are expanded in patients with autoimmune diseases such as lupus, bullous pemphigoid, rheumatoid arthritis (RA) and primary Sjögren's syndrome (pSS) and have been reported to correlate with IL-21 levels, autoantibodies, and disease severity. <sup>26,27,28,29</sup> Furthermore, loss of number and functionality of Tregs has been associated with autoimmune diseases such as SLE and giant cell arteritis, which IL-21 is expected to modulate. <sup>30,31</sup> Thus, neutralization of IL-21 in settings of autoimmunity is expected to impact several cell populations believed to be involved in the pathogenesis of autoimmune disorders including SLE.

BOS161721 selectively binds IL-21 with high affinity to neutralize IL-21, and due to its pleiotropic nature, neutralization of IL-21 is expected to impact several cell populations believed to be involved in the pathogenesis of SLE. Importantly, patients with SLE have elevated IL-21 plasma levels that correlate with the severity of the disease. Recently, genome-wide association studies (GWAS) have provided convincing evidence that the chromosomal 4q 27 region harbors the IL-21 genes and is associated with chronic inflammatory disorders, including SLE.<sup>29</sup>

#### 1.2.2.2 Preclinical Studies

The pharmacokinetics (PK) of BOS161721 were characterized following single-dose intravenous (IV) administration of BOS161721 (0.01 to 30 mg/kg) in male Cynomolgus monkeys or repeat, every 2 weeks IV administration (15 to 100 mg/kg) and subcutaneous (SC) administration (50 mg/kg) in male and female Cynomolgus monkeys. Systemic exposure was approximately dose-proportional within the tested dose range. SC bioavailability was determined to be 64.3%.

Two single-dose (IV) non-good laboratory practice (GLP) studies conducted in Cynomolgus monkeys evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), and immunogenicity of BOS161721. Following a single IV administration (slow bolus), there were no BOS161721-related adverse changes, resulting in a no-observed-adverse-effect-level (NOAEL) value of 30 mg/kg, the highest dose tested among 2 studies.

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) administration for 3 months (a total of 7 doses).




An additional GLP, repeat-dose toxicity study was conducted in Cynomolgus monkeys (4 males and 4 females per dose group) following every 2 weeks (Q2W) administration by SC (10, 30, and 100 mg/kg) injection for a total of 14 doses.

There were no BOS161721-related effects on survival, clinical signs, male body weights, ophthalmologic parameters, electrocardiogram (ECG) findings, clinical pathology, macroscopic observations, organ weights, or microscopic observations.

#### 1.2.2.3 Clinical Studies

BOS161721-01 was a double-blind, Phase 1, single ascending dose (SAD) study to assess the safety, PK, and PD of BOS161721 in healthy subjects. The primary objective of the study was to characterize the safety and tolerability of IV and SC SADs of BOS161721 in an otherwise healthy subject population without concomitant illnesses, immune abnormalities, or concomitant medications. Secondary objectives included characterization of the PK and immunogenicity of BOS161721, and exploratory objectives included the evaluation of the effect of BOS161721 on TDAR to keyhole limpet hemocyanin (KLH) (primary and secondary immunizations) in healthy subjects, the effects of BOS161721 on plasma levels of IL-21 (free and bound), and the evaluation of the effect of BOS161721 on IL-21 gene expression (via gene signature) in blood. This study consisted of 8 cohorts. Subjects were randomized in a 3:1 ratio (BOS161721: placebo) and received either a single dose of BOS161721 (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) or placebo, with safety follow-up. For the first cohort, after the first 2 subjects were dosed (1 active and 1 placebo), there was a minimum gap of 48 hours before the remaining subjects from that cohort were dosed, to allow for an initial review of any emerging safety and tolerability data. For all cohorts, escalation to the next dose was not


Clinical Study Protocol: BOS161721-02


sooner than 8 days after all the subjects in the prior cohort had been dosed and were based on a review of at least 7 days of safety and tolerability data by the Safety Data Monitoring Team (SDMT).

Blood samples were collected at every in-house study visit for BOS161721 concentration determinations. Blood samples were also collected for determination of IL-21 plasma levels (free and total). Safety was assessed based on the occurrence of treatment-emergent AEs, hepatic function abnormality, and acute and delayed hypersensitivity reactions. Other safety variables included ECGs, vital signs (blood pressure [BP], heart rate, and temperature), safety laboratory assessments, blood sampling for ADAs, total IgG and immunoglobulin M (IgM) levels, CD4+ count, and full and targeted physical examinations. Overall, there were no clinically significant findings from this study. Adverse events reported as related to the study drug, particularly infections, were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. There was 1 serious adverse event (SAE; death due to pulmonary embolism) that occurred 127 days after a single administration of 240 mg SC dose of BOS161721. The causality of this single SAE was not attributed to study drug and further information can be found in the Investigator's Brochure. Final PK data from the SAD study demonstrates BOS161721 has a mean t½ ranging from 80 to 87 days for doses of ≥ 30 mg in healthy subjects.

#### 1.2.3 Study Dose Selection

Doses have been selected for the multiple ascending dose (MAD) Phase 1b portion based on a 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01); the SDMT reviewed the blinded safety data from subjects for each dose cohort (8 cohorts, evaluating 1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg), along with the accumulated safety and available PK/PD data from all subjects in the previous dose cohorts, to make a decision on whether to proceed to the next higher dose level, repeat a dose level, or stop dose escalation. Overall, there were no clinically significant safety or tolerability findings from this study.

Based on the Day-90 interim cut of the PK and biomarker data in the BOS161721-01 study, the recommended doses for evaluation in the MAD portion of this study are 20, 60, and 120 mg SC monthly. This dose recommendation is supported by evidence of linear PK with BOS161721 resulting in a median first time to maximum concentration (T<sub>max</sub>) of 6 days and an apparent terminal half-life of 44 days. Furthermore, pSTAT3 suppression, a marker of IL-21 target engagement, follows a similar time course of the mAb levels, with maximal and sustained suppression apparent with doses greater than 30 mg SC (Figure 1).


pSTAT3 cmin percent pSTAT3+ lymphocytes, stimulated) 60 pSTAT3 cmin Route IV · SC 20 100 0 50 150 200 250 Dose (mg)

Figure 1. Individual pSTAT3 C<sub>min</sub> Levels Versus Dose

IV = intravenous, pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SC = subcutaneous

All doses selected for the MAD portion are projected not to exceed the mean exposure of that achieved following the highest single dose of 240 mg SC administered in the Phase 1 SAD study. Cohort 1 will include randomized treatment to the 20 mg dose. Based on the staggered study design, the data monitoring committee (DMC) will perform a scheduled review of safety data and sequentially consider dose escalation for Cohorts 2 and 3. In addition, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the proof of concept (POC) Phase 2 portion. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD portion (see Section 3.1.2.1 for the chosen POC dose and justification).

#### 1.2.4 Risk-Benefit Assessment

The available preclinical data on BOS161721, the findings in clinical study BOS161721-01, and existing clinical information on IL-21 inhibitors suggest that the present clinical study has an acceptable risk-benefit ratio. In this study, the risk-benefit assessment of BOS161721 in adult patients with moderately to severely active SLE will be ongoing, with step-wise evaluations during the staggered MAD portion. The DMC used in this study is charged with assessing such actions in light of an acceptable benefit-risk profile for BOS161721 as an anti-IL-21 mAb.


Formal DMC monitoring meetings will occur as described in the DMC Charter. Two weeks after Cohort 1 has received a second dose of study drug, the DMC will evaluate the safety and tolerability data from Cohort 1 to determine the recommended dose for Cohort 2. Two weeks after 8 patients in Cohort 2 receive a second dose, the DMC will determine if dose escalation to Cohort 3 can proceed. Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 during the MAD part of study. Thereafter, DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter. With the agreement of the DMC and sponsor, this schedule may be modified depending on the rate of patient accrual. Additional details can be found in the DMC Charter.

The benefit of participation for all patients in this study is close monitoring of their medical condition and safety of their treatment. Those randomized to the active treatment arm may potentially experience improvement in their SLE disease. Those randomized to the placebo (in combination with standard of care) arm are not expected to obtain any additional benefit, beyond those of their background treatment, though close monitoring of their medical condition and safety may itself be associated with improving their SLE.

#### 1.2.5 Potential Risks

Potential risks based on the mechanism of action of BOS161721 include infections, risks associated with the administration of any foreign protein or biologic agent, including injection site reaction, anaphylaxis, serious allergic reaction, and development of ADAs. ADAs could result in immune complex disease (with manifestations such as arthralgias, serum-sickness, and vasculitis), or altered BOS161721 levels or activity. Further details can be found in the current Investigator's Brochure (IB) for BOS161721, which contains comprehensive toxicology, preclinical and clinical information on BOS161721.

Two investigational drug products are considered to be in the same pharmacological class as BOS161721 based on interruption of signaling through the IL-21 signaling pathway. No potential risk generalizable across the class has been observed with these investigational products. Based on the clinical Phase 1 SAD study (BOS161721-01), AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc.), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs.

The majority of IgG elimination occurs via intracellular catabolism, following fluid-phase or receptor-mediated endocytosis. This type of endocytosis and elimination is a form of target-mediated disposition where the interaction of the drug and its pharmacological target (eg, a target receptor) serves as a significant contributor to the kinetics of antibody distribution and elimination. Renal elimination, which is a primary pathway of clearance of small-molecule drugs, is relatively unimportant for IgG, as its large size prevents efficient filtration through the glomerulus. Secretion into the bile is an important pathway of elimination of IgA antibodies, but


Clinical Study Protocol: BOS161721-02


this route is not a significant contributor to the elimination of IgG antibodies. Thus, risk to renal and hepatic systems due to metabolism of BOS161721 is low.<sup>33</sup>

## 1.2.5.1 Anaphylaxis and Serious Allergic Reactions

As with the administration of any foreign protein and/or other biological agents, acute hypersensitivity reactions, including acute anaphylactic/hypersensitivity, severe allergic, and anaphylactoid reactions may follow infusion of mAbs and can be caused by various mechanisms. These acute hypersensitivity reactions may be severe and result in death.

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria,<sup>34</sup> and are discussed in Section 6.2.2.6.1.

Based on the Phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed.

Patients with a known history of allergy or severe hypersensitivity reaction to any component of BOS161721 formulation or patients with a history of anaphylaxis to any other biological therapy such as mAbs will be excluded from studies with BOS161721. In addition, appropriate drugs and medical equipment to treat acute hypotensive, bronchoconstrictive, or anaphylactic reactions will be immediately available at the unit and study personnel will be trained to recognize and treat these reactions.

#### 1.2.5.2 Injection Site Reactions

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC for 3 months (a total of 7 doses). There were no injection site reactions in animals dosed subcutaneously. Further, there were no reports of injection site reactions in the 26-week GLP toxicology study in Cynomolgus monkeys.

Based on the Phase 1 SAD study (BOS161721-01), incidence of injection site reactions in subjects who received BOS161721 was similar to placebo.

Patients will be monitored for local injection site reactions in this study. See Section 6.2.7.

#### 1.2.5.3 Immune Complex Disease

The potential risk of immune complex disease for BOS161721 is theoretical, based on the known risks associated with mAbs. The administration of a mAb can result in the formation of ADAs. Administration of the mAb in the presence of ADA may result in the formation of circulating antibody-antigen complexes potentially resulting in altered BOS161721 levels or activity or deposition of the complexes in microvasculature. Complement is frequently involved in the latter setting, and the breakdown products of complement attract polymorphonuclear leukocytes to the site of deposition where they can provoke local tissue damage through specific or nonspecific release of enzymes. Two of the more common end-organ targets are the blood vessels (vasculitis) and kidney (nephritis). These clinical manifestations represent immune complex disease or Type III hypersensitivity. Although BOS161721 is a humanized mAb,


Clinical Study Protocol: BOS161721-02


ADAs may develop; however, the likelihood of occurrence of immune complex disease with BOS161721 is low. The findings of immune complex disease are typically reversible when mAb administration stops and the antibody-antigen complexes are cleared from the body.

Based on the Phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed.

#### 1.2.5.4 Infections

BOS161721 is expected to diminish the activity of T-cell, B-cell and NK-cell lines. Like other medications modulating immune response, BOS161721 may increase the potential risk for infection, including serious infections. IL-21 produced by CD4+ Th cells is required to sustain the anti-viral function of CD8+ T-cells against chronic viral infections. Nonclinical evidence suggests that the risk of chronic viral infection recurrence or increased severity may occur with IL-21 inhibition.<sup>35</sup>

These conditions will be fully characterized with clinical descriptions and routine laboratory and/or specialty testing and treated where indicated with appropriate local standard of care.

Patients with a history of opportunistic infection, including recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years, or any other underlying pathology predisposing to serious infection, are excluded from studies with BOS161721 (for further details please refer to the current IB for BOS161721).

Patients will be assessed for hepatitis B, and C, and HIV-1/2 combination, at screening.

## Cryptosporidium Infection

Cryptosporidium infection was noted in patients with an IL-21 receptor loss-of-function gene mutation and similar findings of cryptosporidium infection have been observed in immunosuppressed liver transplant and human immunodeficiency virus patients. Since BOS161721 is expected to diminish the immunosurveillance activity of T-cell, B-cell, and NK-cell lines, a similar risk is biologically plausible with prolonged exposure to BOS161721.

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells,<sup>37</sup> patients with a CD4+ count < 500 cell/mm³ were excluded from the Phase 1 SAD study (BOS161721-01), and CD4 + < 350 cells/mm³ will be excluded from the MAD/POC parts of the study. Patients exposed to investigational product who develop diarrhea during the course of the study should immediately undergo an assessment for opportunistic infection including stool for ova and parasites and stool examination for cryptosporidium. Positive cryptosporidium in stool sample at screening is an exclusion. Treatment by the investigator where indicated should be guided by findings and be consistent with local standard of care.

Based on the Phase 1 SAD study (BOS161721-01), infections in subjects who received BOS161721 was not observed.


## 1.2.5.5 Malignancy

The stimulatory effect of IL-21 on NK cells and CD8+ T-cells suggests the cytokine may have anti-tumor activity. Nonclinical studies have demonstrated significant anti-tumor effects of IL-21 in a number of tumor models. IL-21 therapy of human metastatic melanoma and renal cell carcinoma has demonstrated POC with significant increases in levels of perforin, granzyme B, and interferon gamma (IFN $\gamma$ ) expression in CD8+ T-cells and NK T-cells. Clinical response has been limited in these generally unmanageable diseases.

The impact of treatment with anti-IL-21 therapy on the development or growth of malignancies is not known; however, as with other immunomodulatory biologic agents, treatment with BOS161721 may result in an increase in the risk of malignancies. NK cell suppression by IL-21 neutralization may represent a biological mechanism for a potential risk for malignancy. Patients with a history or current diagnosis of cancer within the past 5 years, with the exception of non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy, are excluded from the study.

Based on the Phase 1 SAD study (BOS161721-01), malignancy in subjects who received BOS161721 was not observed.

### **1.2.5.6** Hepatic Function Abnormality

There is no substantial evidence suggesting BOS161721 is associated with liver function abnormality. However, as a precaution, patients with a history of abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST >  $2 \times \text{upper limit of normal [ULN]}$ ; total bilirubin >  $1.5 \times \text{[ULN]}$  and judged by the investigator to be clinically significant) were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from this trial. Patients with a positive hepatitis B or C test or a history of alcohol dependence will also be excluded.

Based on the Phase 1 SAD study (BOS161721-01), hepatic function abnormality in subjects who received BOS161721 was not observed.

#### 1.2.5.7 Failure of Vaccination

IL-21 is a key cytokine in development of B-cells into immunoglobulin-secreting plasma cells. Abnormal signaling through the IL-21R/Janus Kinase (JAK)3/signal transducer and activator of transcription (STAT3) pathway leads to defective humoral immune responses to both T-dependent and T-independent antigens and impairs the establishment of long-lasting B-cell memory. Abnormal signaling through the pathway has been related to decreased specific antibody responses following vaccination, and to increased susceptibility to encapsulated bacterial infections.<sup>38</sup>

The effect of BOS161721 was evaluated in *in vivo* single dose studies in Cynomolgus monkey in which the animals received vaccination to T-cell dependent KLH antigen to stimulate a TDAR. These *in vivo* studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen in a dose-dependent fashion; however,


BOS161721 administration did not affect anti-tetanus toxoid antibody data for IgM, IgG, IgG1, or immunoglobulin E (IgE) during the dosing phase in the same study.

## 1.2.5.8 Potential for Drug-Drug Interactions

Drug-drug interactions were not evaluated in the Phase 1 SAD study (BOS161721-01), which included only healthy adult subjects. Use of prescription medications (with the exceptions of oral contraceptives), and over-the-counter (OTC) treatments including herbal supplements such as St John's Wort (except multivitamins), in the 2 weeks prior to screening was prohibited in the SAD study.

See Section 4.5 for other specific exclusion criteria which support lowered risk of interactions, and Section 4.6.1 for corticosteroid (CS) dosing. In addition, Section 1.2.5.6 describes considerations for hepatic function for this study.

## 1.2.5.9 Potential Risk to Fetal Development

No data on preclinical reproductive toxicity are available at the time of this study.

#### 2 STUDY OBJECTIVES AND ENDPOINTS

This trial has separate objectives and endpoints for the MAD Phase 1b and POC Phase 2 portions of the study. The primary, secondary, and exploratory objectives for each phase, as applicable, are described below with their corresponding endpoints.

# 2.1 Phase 1b Multiple Ascending Dose

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optima dose. | Safety Endpoints Incidence and severity of AEs and SAEs, related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness Injection site reactions Columbia Suicide Severity Rating Scale (C-SSRS) 12-lead ECGs parameter results at each visit and change from baseline Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline Clinical laboratory results and change from baseline Physical examinations changes from baseline ADAs Study drug exposure/compliance |
| Secondary | |
| To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PI effects in patients with moderately to | <ul> <li>Pharmacokinetic Endpoints</li> <li>BOS161721 concentration by visit and time point</li> <li>Maximum observed concentration (C<sub>max</sub>), T<sub>max</sub>, area under the concentration-time curve (AUC), terminal elimination</li> </ul> |


Protocol Date and Version: 23 January 2019; V5.0 severely active SLE. half-life (t<sub>1/2</sub>), systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>) Pharmacodynamic Endpoints Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit **Exploratory** CCI


Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 23 January 2019; V5.0

# Phase 2 Proof of Concept

| DINTS |
|---|
| Efficacy Endpoint e proportion of patients with a SRI-4 response at y 210 (see Section 6.3.4.1) |
| DOS DE LES |
| ary Efficacy Endpoints e proportion of patients with: SRI-4 response at each visit SRI-5 and SRI-6 response at each visit (Section 6.3.4.2) a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210 new BILAG A flare or > 1 BILAG B flares relative to baseline through Day 210 PGA worsening a BICLA response a CLASI response medication failures sults and changes from baseline in: CLASI swollen and tender joints ACR-28 SLEDAI-2K SLICC/ACR damage index ne to medication failure ration of longest SRI-4 response ne to first SRI-4 response ne to BILAG A flare or > 1 BILAG B flare compared to eline through Day 210 |
| 7 1 ' , |
| Endpoints idence and severity of adverse events (AEs) and serious verse events (SAEs), related AEs, AEs leading to study g discontinuation, AEs by severity and relatedness ection site reactions SSRS lead ECGs parameter results at each visit and change m baseline al signs (blood pressure [BP], heart rate, and apperature) parameter results at each visit and change m baseline inical laboratory results and change from baseline visical examinations changes from baseline |
| 1 |

# Exploratory


Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 23 January 2019; V5.0



#### 3 STUDY PLAN

# 3.1 Study Design

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, eligible patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly.

The trial will consist of 2 double-blinded portions: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

SLE disease activity assessment data will be centrally reviewed by medical monitor and sponsor to ensure the scores are clinically meaningful and compliant with specific definition. The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease activity. Further details on the content and methods of data reports by the medical monitor and sponsor will be outlined in the Medical Data Review Plan along with the processes and procedures that will be followed.

## 3.1.1 Multiple Ascending Dose Phase 1b

The MAD portion will consist of 3 cohorts:

• Cohort 1 (20 mg SC) will include 6 patients


Clinical Study Protocol: BOS161721-02


o 5 patients will receive BOS161721 (active group) and 1 patient will receive placebo (placebo group)

- Cohorts 2 (60 mg SC) and 3 (120 mg SC) will include 12 patients each
  - o 9 patients in the active group and 3 in the placebo group

Doses selected for each of the 3 cohorts is based on a 90-day safety, tolerability, PK and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. All doses selected for the MAD part of the study are projected not to exceed the mean exposure of that achieved in the SAD study.

#### 3.1.1.1 Dose Escalation for the MAD Portion

The MAD portion of the study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after the DMC evaluation of the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after the DMC evaluation of the safety and tolerability data from Cohorts 1 and 2. Each cohort will continue at their assigned dose level through their respective 6-month treatment periods (See Study Schematic, Section 3.1). If patients discontinue the study in a cohort prior to adequate safety follow-up, he/she may be replaced.

Criteria for dose escalation are further described in the DMC Charter. See Section 3.1.1.2 for additional details about DLTs.

#### 3.1.1.2 Dose Limiting Toxicity (DLT)

Severity of adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs occurring after study drug administration, which are attributable to the study drug, will be considered DLTs:

#### **Hematologic:**

- Grade 4 neutropenia
- Grade 3 neutropenic infection
- Grade 3 thrombocytopenia with bleeding
- Grade 4 thrombocytopenia

#### **Non-Hematologic:**

• Grade 3 or above toxicities, persisting after optimal treatment with standard medical therapy (eg, anti-emetics, anti-diarrheals)


Clinical Study Protocol: BOS161721-02


• Drug-induced liver injury ([DILI], Hy's Law), as defined in Section 6.2.2.6.3

Investigators should always manage their patients according to their medical judgment which may include interruption of study drug based on the particular clinical circumstances.

#### 3.1.1.3 DMC Recommendations

During scheduled meetings, the DMC will review relevant study data for safety or benefit-risk concern. During the MAD part of the study, the DMC may provide the following recommendations to the sponsor:

- Expanding a cohort at a specific dosing level, or repeating a lower dose in a subsequent cohort
- Continuing a dose level for a given cohort
- Escalating a dose level for a subsequent cohort
- Termination of current or previous cohort(s)

Further dosing in a given cohort will be halted if 2 or more DLTs are identified intra- and inter-patients dosed. For the POC portion, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC Phase 2 part of the study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD portion. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available 30 days after the last patient from Cohort 3 receives the third dose. Details are provided in the DMC Charter.

## **3.1.2 POC Phase 2**

#### 3.1.2.1 BOS161721 POC Dose Selection and Justification

The dose for the POC portion of the study is 120 mg administered SC monthly (a total of 7 doses). The rationale for the BOS161721-02 Phase 2 POC dose selection was based on cumulative safety, tolerability, immunogenicity, PK, and PD data available from an interim analysis (IA) performed during the MAD Phase 1b portion of the trial.

The data cut-off for this IA occurred on CCl and and included all 6 patients and 7 doses from Cohort 1 (20 mg), 12 patients and 6 doses from Cohort 2 (60 mg), and 12 patients and 4 doses from Cohort 3 (120 mg).

The safety analysis focused on incidence and severity of all AEs, SAEs, and pre-determined adverse events of special interest (see Section 6.2.2.6). The DMC and designated unblinded Boston Pharmaceuticals team met on CCI and did not identify any untoward safety signals at any BOS161721 dose levels.


Clinical Study Protocol: BOS161721-02


Because there were no safety, tolerability, or immunogenicity trends observed at the time of the IA, the Phase 2 POC dose selection was made based on available PK and PD data. pSTAT3 levels were assessed as the primary PD biomarker of IL-21R signaling levels. This is because IL-21R signaling, upon IL-21 binding, initially involves phosphorylation of JAK1/JAK3 which dissociate from the receptor complex, and phosphorylate STAT3 which translocates to the nucleus and drives IL-21-regulated gene expression.

The 120 mg dose will be communicated to site investigators participating in the POC Phase 2 portion, and to Institutional Review Boards (IRBs) and the Independent Ethics Committee (IEC).

## 3.1.2.2 POC Study Design

For the POC part of the study, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio.

As in the MAD part of the study, each patient in the POC portion may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Section 3.4).

DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.

# 3.2 Randomization and Blinding

This is a randomized, double-blind study.

Patients meeting all inclusion and exclusion criteria will be centrally randomized to either placebo or BOS161721 using an IWRS according to a randomization list generated by an independent, non-study statistician. Randomization will be performed separately for each study portion and separately for each cohort in the Phase 1b and 2 portions as follows:

| Phase/Cohort | Number of Patients | Randomization Ratio BOS161721:Placebo |
|---|---|---|
| Phase 1b/Cohort 1 | 6 | 5:1 |
| Phase 1b/Cohort 2 | 12 | 3:1 |
| Phase 1b/Cohort 3 | 12 | 3:1 |
| Phase 2 | 156* | 2:1 |

<sup>\*</sup>Additional patients may be enrolled to ensure sufficient numbers of patients are in the full analysis set (FAS).

Eligible patients will be assigned to the study portion which is active at time of enrollment. Similarly, patients in the Phase 1b MAD will be assigned to the cohort which is active. Each patient will be assigned a unique randomization number which will not be reused.

All patients, investigators, and study team participants will be blinded to treatment assignment. An independent biostatistician not otherwise involved on the study will be unblinded and prepare materials for the IA, ad hoc analyses as needed, and the DMC safety reviews. The DMC will


Clinical Study Protocol: BOS161721-02


review unblinded data during safety reviews and the IA. A limited team at Boston Pharmaceuticals will review unblinded results from the Phase 1b MAD portion during the IA to determine the dose that will be used for the Phase 2 POC portion of the study. Details regarding maintenance of the blinding and content of data reviews will be described in the DMC charter or related study documentation.


Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 23 January 2019; V5.0

## 3.3 Study Schematic

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2



A = active drug (BOS161721); P = placebo


Clinical Study Protocol: BOS161721-02


# 3.4 Schedule of Assessments

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | Treatment Period Follow-Up | | | | | | | | | | | | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| GENERAL ASSESS | MENTS | | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| SLICC Criteria for<br>SLE | X | | | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>c</sup> | | X | | | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | | X | | X | X | X | X | X | | | | | |
| SAFETY ASSESSM | ENTS | | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | | | |
| Chest x-ray <sup>d</sup> | X | | | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>e</sup> | X | X | | | X | | | X | | | | | | | | X |
| Injection site reaction assessment | | X <sup>f</sup> | X | | X | | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | | X | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>g</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESS | SMENTS | | | | | | | | | | | | | | | |
| BILAG-2004 Index | X | X | | | X | | X | X | X | X | X | | | X | X | X |


Clinical Study Protocol: BOS161721-02


Table 1. Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | Treatment Period Follow-Up | | | | | | | | | | | | Safety Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| SLEDAI-2Kh | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| PGA of disease activity | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CCI | 71 | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLICC/ACR | | | | | | | | | | | | | | | | |
| Damage Index | | X | | | | | | | | | X | | | | | |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| LABORATORY ASS | SESSMEN | TS | | | | | | | | | | | | | | |
| CD4+ count | X | X | | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments (hematology and | | | | | | | | | | | | | | | | |
| clinical chemistry) <sup>i</sup> | X | X | | | X | X | X | X | X | X | X | | | X | X | X |
| Coomb's test direct | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | | X | X | X | | X | | | X | | | | | |
| Plasma CC | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Plasma CCI & | | X | | X | X | | X | X | | | X | | | | | |
| Whole blood for | | | | | | | | | | | | | | | | |
| leukocyte | | | | | | | | | | | | | | | | |
| immunophenotype | | X | | X | X | | X | X | | | X | | | | | |
| ADA <sup>k</sup> | | X | | X | X | | X | X | | | X | | | | | X |
| nAb <sup>l</sup> | | | | | | | | X | | | X | | | | | |
| pSTAT3 <sup>m</sup> | | X | | | X | X | X | X | | | | | | | | |
| CCI | | X | | X | | | | X | | | X | | | | | X |
| CCI | | X | | | | | | | | | | | | | | |


Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 23 January 2019; V5.0

**Schedule of Assessments - Phase 1b - Multiple Ascending Dose** Table 1.

| | Screena | Enroll | | Treatment Period Follow-Up | | | | | | | | | | | | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| CCI | X | X | | | X | | X | X | X | X | X | | | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> |
| CRP | X | | | | | | | X | | | | | | | | X |
| Serum pregnancy<br>test (women) | X | | | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>o</sup> | | X | | | X | | X | X | X | X | X | | | | | X |
| TB test<br>(QuantiFERON-TB<br>Gold In-Tube) <sup>d</sup> | X | | | | | | | | | | | | | | | |
| Serology (hepatitis<br>B and C, HIV-1/2<br>combination) | X | | | | | | | | | | | | | | | |
| Stool sample <sup>p</sup> | X | | | | | | | | | | | | | | | |
| Spot urine for protein/creatinine ratio | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | | X | | X | X | X | X | X | | | X | X | X |


Clinical Study Protocol: BOS161721-02


**Table 1.** Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Tre | eatment | Period | Follow- | Up | | | | Safet | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | $(\pm 3)$ | $(\pm 3)$ | $(\pm 3)$ | $(\pm 3)$ | $(\pm 3)$ | $(\pm 3)$ | (± 3) | $(\pm 3)$ | $(\pm 3)$ | $(\pm 3)$ | $(\pm 3)$ | (± 3) | $(\pm 3)$ |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| PK Labs | | | | | | | | | | | | | | | | |
| Predose | | X | | | X | | X | X | X | X | X | | | | | |
| Predose PK<br>Window | | 60m | | | ± 3d | | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | | | | | |
| Postdose | | Xq | X | X | Xq | | ± 3u | ± 3 <b>u</b> | ± 3 <b>u</b> | ± 3 <b>u</b> | X <sup>q</sup> | X | X | X | X | X |
| Postdose PK<br>Window | | 4h ± 30m<br>8h ± 45m<br>24h ± 60m | ± 1d | ± 3d | 4h ± 30m<br>8h ± 45m<br>24h ± 60m | | | | | | 4h ± 30m<br>8h ± 45m<br>24h ± 60m | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CC ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; d = day; ECG = electrocardiogram; FSH = follicle stimulating hormone; h = hour; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; m = minute; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SAE = serious adverse event; SC = subcutaneous; CC | SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics;

<sup>a</sup> Screening assessments will be performed over more than 1 visit.

Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 4.6.1 for further details.

; TB = tuberculosis; TDAR = T-cell dependent antigen response.

- <sup>c</sup> Randomization should occur after patient eligibility has been confirmed by central eligibility review.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- <sup>e</sup> ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed at 2 hours postdose.
- yital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, 187, and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.


Clinical Study Protocol: BOS161721-02


 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | Treatment Period Follow-Up | | | | | | | | | | | | fety Follow-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 7 15 30 44 60 90 120 150 180 187 195 | | | | | | | | | | | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | - | 11 | 12 | 13 |

- SLEDAI-2K should be done before randomization and dosing on Day 0 as SLEDAI-2K < 6 is exclusionary.
- <sup>1</sup> Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.
- When clinically indicated for hemolytic anemia.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed (analyzed) if the patient had a positive ADA on Day 90.
- <sup>1</sup> nAb is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90.
- m Predose (trough) samples only.
- <sup>n</sup> Only CCl collected during safety follow-up visits.
- <sup>o</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- P Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- <sup>q</sup> Postdose samples will be collected at 4, 8, and 24 hours after study drug administration on Days 0, 30, and 180.


Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 23 January 2019; V5.0

Schedule of Assessments - Phase 2 Proof of Concept (POC) Table 2.

| | Screena | Enroll | | | | Safe | Safety Follow-Up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | 2337 032 | 15 | 30 | 60 | reatment<br>90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| GENERAL ASSESSMENTS | · | | | | | • | | • | | | • | | • | |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| SLICC Criteria for SLE | X | | | | | | | | | | | | | |
| Concomitant medication <sup>c</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>d</sup> | | X | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | X | X | X | X | X | X | | | | | |
| SAFETY ASSESSMENTS | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | |
| Chest x-ray <sup>e</sup> | X | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>f</sup> | X | X | | X | | X | | | | | | | | X |
| Injection site reaction | | | | | | | | | | | | | | |
| assessment | | Xg | | X | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and | 77 | 77 | 37 | *** | 37 | 37 | 37 | *** | *** | | | 37 | 37 | 7.7 |
| temperature)h | X | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESSMENTS | T 77 | 77 | | | 37 | | | | | ı | 1 | | | 77 |
| BILAG-2004 Index | X | X | | X | X | X | X | X | X | | | X | X | X |
| SLEDAI-2K | X | Xi | | X | X | X | X | X | X | | | X | X | X |
| PGA | X | X | | X | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | X | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | X | X | X | X | X | X | | | X | X | X |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |


Clinical Study Protocol: BOS161721-02


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | Treatment Period Follow-up | | | | | | | | | | | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | - | | 10 | 11 | 12 |
| SLICC/ACR Damage Index | | X | | | | | | | X | | | | | |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |
| LABORATORY ASSESSMENT | S | | | | | | | | | | | | | |
| CD4+ count | X | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments | | | | | | | | | | | | | | |
| (hematology and clinical | | | | | | | | | | | | | | |
| chemistry) <sup>j</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Coomb's test direct <sup>k</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | X | X | | X | | | X | | | | | |
| Plasma CC | X | X | | X | X | X | X | X | X | | | X | X | X |
| Plasma CCI & CCI | | X | X | X | | X | | | X | | | | | |
| Whole blood for leukocyte | | | | | | | | | | | | | | |
| immunophenotype | | X | X | X | | X | | | X | | | | | |
| ADA <sup>1</sup> | | X | X | X | X | X | | | X | | | | | X |
| nAb <sup>m</sup> | | | | | | X | | | X | | | | | |
| CCI | | X | X | | | X | | | X | | | | | X |
| CCI | | X | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | |
| | X | X | | X | X | X | X | X | X | | | Xn | X <sup>n</sup> | X <sup>n</sup> |
| CRP | X | | | | | X | | | | | | | | X |
| Serum pregnancy test (women) | X | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>o</sup> | | X | | X | X | X | X | X | X | | | | | X |
| TB test (QuantiFERON-TB Gold In-Tube) <sup>e</sup> | X | | | | | | | | | | | | | |
| Serology (hepatitis B and C,<br>HIV-1/2 combination) | X | | | | | | | | | | | | | |


Clinical Study Protocol: BOS161721-02


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | Т | reatmen | t Period | Follow-u | ıp | | | Safet | y Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | to -1 | 0 | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| Stool sample <sup>p</sup> | X | | | | | | | | | | | | | |
| Spot urine for protein/creatinine | | | | | | | | | | | | | | |
| ratio | X | X | | X | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | X | X | X | X | X | X | | | X | X | X |
| PK Labs <sup>b</sup> | | | | | | | | | | | | | | |
| Predose | | X | | X | X | X | X | X | X | | | | | |
| Postdose | | | X | | | | | | | X | X | X | X | X |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CC ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; d = day; ECG = electrocardiogram; CC ; FSH = follicle stimulating hormone; h = hour; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; m = minute; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; SAE = serious adverse event; SC = subcutaneous; CC ; SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; CC ; TB = tuberculosis;

TDAR = T-cell dependent antigen response.

- <sup>a</sup> Screening assessments will be performed over more than 1 visit.
- PK samples will only be collected at the investigational sites that participate in the PK portion of the study. On PK only days (ie, Day 187 and Day 195 when no laboratory assessments are scheduled) samples will be collected at the investigational sites of the selected countries that participate in the PK portion of the study. Patients not participating in PK are not required to return for investigation site visits on Days 187 and 195.
- <sup>c</sup> Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 4.6.1 for further details.
- Randomization should occur after patient eligibility has been confirmed. The actual randomization procedure can be completed on Day -1 after eligibility confirmation or the morning of Day 0 prior to dosing for logistical purposes.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- g Injection site reaction assessments to be performed at 2 hours postdose.
- <sup>h</sup> Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 187 and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.


Clinical Study Protocol: BOS161721-02


 Table 2.
 Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | Treatment Period Follow-up | | | | | Safet | Safety Follow-Up | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 <sup>b</sup> | 195 <sup>b</sup> | 210 | 240 | 270 |
| Days | to -1 | 0 | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ | $(\pm 3)$ | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |

- SLEDAI-2K should be done before randomization and dosing on Day 0 as SLEDAI-2K < 6 is exclusionary.
- Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.
- k When clinically indicated for hemolytic anemia.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed (analyzed) if the patient had a positive ADA on Day 90.
- m Ab is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90.
- n Only CCl collected during safety follow-up visits.
- Our Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- P Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.


## 3.5 End of Study

End of Study (Individual Patient): A patient is considered at the end of study if he/she has withdrawn, prematurely discontinued, or completed all of the study procedures including the last visit.

End of Study (End of trial): The end of the study is defined as the date of the last visit of the last patient in the study globally, or the date of which the last patient withdraws or discontinues if all prior enrolled patients have already completed/withdrawn.

## 4 POPULATION

## 4.1 Participant Recruitment

Advertisements approved by the IRB, and investigator databases, may be used as recruitment procedures for adult men and women with moderately to severely active SLE.

### 4.2 Number of Patients

Approximately 186 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD Phase 1b portion, and approximately 156 additional patients will be randomized in the POC Phase 2 portion. Note that approximately 24 dropouts are assumed.

# 4.3 Patient Screening

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Section 3.4]) for this study must be performed between Day -28 and Day -1.

#### 4.4 Inclusion Criteria

Patients who meet the following criteria will be considered eligible to participate in this clinical study:

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1


immunologic criterion or Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously

- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq 1:80$  via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
  - c. C3 or C4 levels below normal as determined by central lab
- 5. At screening, the SLE Disease Activity Index 2000 (SLEDAI-2K) must be ≥ 6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 7. Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - i. "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis in ≥ 2 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living that has been present on several days cumulatively over the past 30 days, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
      - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):


 Ambulation, toileting, grooming- including bathing and dressing; feeding oneself

- ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in ≥ 1 joint, (observed or throughout history), with some loss of functional range of movements manifested by effects on instrumental ADLs such as:
  - Cooking, driving, using the telephone or computer, shopping, cleaning, etc., and has been present on several days over the last 30 days, and is present at the time of the screening visit

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization) (see APPENDIX 3)
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

#### 4.5 Exclusion Criteria

Patients presenting with any of the following will not be included in this study:

1. Drug-induced SLE, rather than "idiopathic" SLE


2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic sclerosis, or vasculitis not related to SLE)

- a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed.
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study. (See Section 4.6 for prohibited concomitant medication)
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening


- 15. CD4+ count < 350/μL at screening
- 16. Platelets < 50,000/mm<sup>3</sup> (50  $\times$  10<sup>9</sup>/L) or < 35,000/ mm<sup>3</sup> (35  $\times$  10<sup>9</sup>/L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation<sup>39</sup>:

GFR = ([1 for male] or [0.85 for female]) 
$$\times$$
 (140 – Age)  $\times$  BW / (72  $\times$  Creatinine)

- 20. Serum ALT and/or serum AST  $> 2 \times ULN$  at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK)  $> 3.0 \times$  ULN at screening, unless it is related to lupus myositis
- 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (eg, IgG protein) or molecules made of components of monoclonal antibodies
- 25. History substance and/or alcohol abuse or dependence within the past 1 year, at the investigator's judgment
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision)
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4 or 5 on the C-SSRS
- 31. Current or pending incarceration


Clinical Study Protocol: BOS161721-02


32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness

#### 4.6 Concomitant Medications

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Patients should stay on stable regimen of other concomitant medications for the treatment of SLE (eg, analgesics, NSAIDs, statins, ACE inhibitors/ARBs and other antihypertensive drugs), unless changes in these treatments are clinically indicated. Use of any other drugs for non-SLE conditions, including over-the-counter medications and herbal preparations, should remain stable unless change or addition is clinically necessary. Discussion with the medical monitor prior to initiation of new medication is strongly recommended. Any concomitant therapies must be recorded on the eCRF. Prior and concomitant medication use will be recorded for the 30 days prior to screening until the last follow-up visit. In addition, historical treatment for SLE (including immunosuppressant, anti-malarial, corticosteroid, and/or biologic agent) will be recorded for the 48 weeks prior to screening in the eCRF.

#### 4.6.1 Corticosteroid

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day).

Tapering of steroids during the course of the study will be highly encouraged and should be evaluated at the protocol permitted visits (Day 0 through Day 60 and Day 120 through Day 150). Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant due to the endpoint evaluations occurring at Day 120 and Day 210.

- Once a patient has received the first dose of study drug (after Day 0), prednisone (or prednisone equivalent) dose is highly encouraged to continue tapering down as appropriate. The investigator should evaluate the prednisone dose at each visit and make the decision, within the protocol allowed windows.
  - Exception: Between Day 60 and Day 120, and between Day 150 and Day 210 (ie, within 60 days of primary and secondary endpoint assessments), oral CS doses must be held constant.

After Day 0 (first dose of study drug), a maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed between Day 0 and Day 60, according to the following:

• The oral CS dose is allowed to increase to  $\leq 40$  mg/day of prednisone or equivalent, which must be tapered down to  $\leq 10$  mg/day within 2 weeks of initiation of the "burst"


O Alternatively, a single intramuscular (IM) dose of methylprednisolone (40 mg or equivalent) is permitted

o No increase of oral CS above baseline is permitted beyond Day 60

Treatment with inhalational CS therapy (eg, for asthma), or by any other route, but systemic administration, is allowed.

Treatment with intra-articular or intravenous CS is prohibited during the course of the study.

#### 4.6.2 Other Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in APPENDIX 4. Medications taken within 30 days prior to screening must be recorded on the eCRF.

- 1. Prior exposure to BOS161721
- 2. Patients who have received treatment with anti-CD20 monoclonal antibodies within 24 weeks of screening; recovery of B cells (CD19+) must be documented (record absolute number of CD19+ B cells)
- 3. Patients who have received treatment with cyclophosphamide within the 24 weeks prior to screening
- 4. Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria within 4 weeks for oral use or 8 weeks for topical use of screening
- 5. Patients who are currently receiving or are scheduled to receive plasmapheresis or lymphapheresis therapy, or have received such therapy within 24 weeks prior to screening
- 6. Patients who have received any live vaccines within 30 days of screening. Note: Furthermore, live vaccines should not be used during the course of the study and within the 2 months following last dose. Other inactivated vaccines such as tetanus, etc., may be used according to local guidelines during treatment period
- 7. Patients who are scheduled or anticipated to have elective surgery during the course of the study
- 8. Initiation of new immunosuppressant or anti-malarial agent is not permitted. Note: Dose reduction or replacement may be allowed due to intolerability or shortage for patients on a stable dose prior to study initiation

# 4.7 Women of Childbearing Potential

WOCBP is defined as any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) and is not postmenopausal.

See Section 4.7.2 for detailed information regarding contraceptive requirements for WOCBP.


## **4.7.1 Determination of Menopause**

Menopause is defined as at least 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes. Women under the age of 55 years must have a documented serum FSH level > 40 mIU/mL at screening to confirm menopause.

### 4.7.2 Contraception

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks, due to the mean terminal ½ life of the study drug.

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks, due to the mean terminal ½ life of the study drug.

Investigators shall counsel WOCBP and men who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and men who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, patients must agree to the use of 1 method of highly effective contraception from the following:

- Male condoms with spermicide
- Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as 1 of the acceptable methods of contraception since they will not be receiving study drug.
- IUDs, such as ParaGard®
- Vasectomy
- Complete abstinence, defined as complete avoidance of heterosexual intercourse, is an acceptable form of contraception. Women who are abstinent while participating in the study must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the patient chooses to forego complete abstinence.

Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing.

#### 4.8 Deviation from Inclusion/Exclusion Criteria

Deviation from the inclusion or exclusion criteria will not be allowed. If deviation of inclusion/exclusion criteria is discovered after randomization, the investigator should contact the medical monitor for discussion. A decision will be made whether to allow a patient to continue or withdrawal from the study medication.


Clinical Study Protocol: BOS161721-02


See Section 6.8 for additional details.

### 4.8.1 Patient Withdrawal and Replacement

See Section 5.5 for reasons for removal from the trial. Withdrawn patients may be replaced during the MAD part of the study after discussion between the principal investigator or designee and sponsor.

### 5 STUDY PROCEDURES

Refer to the eCRF completion guidelines for data collection requirements and documentation of study assessments/procedures.

## 5.1 Screening

Screening will be the same for both the MAD and POC portions of the study.

Screening will take place from Day -28 to Day -1, and assessments may be performed over more than 1 visit. Confirmation that the most current IRB/IEC approved informed consent form (ICF) has been signed must occur before any study-specific screening procedures are performed. Procedures that are part of standard of care are not considered study-specific procedures and may be performed prior to informed consent and used to determine eligibility.

All screened patients will be assigned a unique screening number. The screening number will include a 3-digit site number and a 4-digit sequential number to identify patients from the time of screening. Only eligible patients who are confirmed by central review as meeting the inclusion/exclusion criteria, listed in Section 4.4 and Section 4.5 respectively, will be enrolled in the study. Screened patients who drop out of the clinical study before randomization will be recorded as screen failures. If rescreening occurs, the site will assign a new screening number.

Specific procedures at the screening visit will include:

- Medical history documentation
- Review of inclusion and exclusion criteria
  - o Patient medical records must contain documentation of SLE diagnosis
  - o C-SSRS
- Concomitant medication documentation
- Demographics
- Full physical examination
- Vital signs
- Chest x-ray (a prior x-ray can be used if taken within 12 weeks of screening date)
- Laboratory evaluations (non-fasting):
  - o Hematology and clinical chemistry
  - o Serology (Hepatitis B and C; HIV-1/2 combination)
  - o TB test


Clinical Study Protocol: BOS161721-02


- o CRP
- o Direct Coomb's test (if indicated for hemolytic anemia)
- o CD4+ count, total IgG and IgM levels, plasma CC , CCl
- Serum pregnancy test (WOCBP)
- o FSH (postmenopausal women under age 55 years)
- o Spot urine for protein/creatinine ratio
- o Urinalysis
- Stool sample
- 12-lead ECG
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, Physician's Global Assessment (PGA) of disease activity

Screening procedures are listed in the Schedule of Assessments (Section 3.4), and details are provided in Section 6.

## **5.1.1** Retesting During Screening Period

A single retesting of laboratory parameters and/or other assessments during the screening period is permitted (in addition to any parameters that require a confirmatory value) only if:

- medically indicated
- there is evidence a laboratory sample was mislabeled, indeterminate, inadequately processed, and/or deteriorated in transit to the central laboratory

Any new result will override the previous result (ie, the most current result prior to randomization) and is the value by which study inclusion/exclusion will be assessed, as it represents the patient's most current clinical state. This will also apply to patients who are being rescreened.

## 5.2 Enrollment/Randomization and Day 0 Treatment

Randomization should occur after patient eligibility for enrollment has been confirmed by the central eligibility review.

Prior to randomization, the study site should confirm that the patient still meets inclusion/exclusion criteria (especially SLE disease activity and treatment). The site will obtain a randomization number when registering the patient in IWRS. All patients will receive BOS161721 or placebo according to the kit number assigned by the IWRS randomization scheme.

After randomization, procedures include:

- PROs: CC
- C-SSRS
- Laboratory evaluations (fasting):


- Hematology and clinical chemistry
- o Direct Coomb's test (if indicated for hemolytic anemia)
- o CD4+ count, total IgG and IgM levels, plasma CCl and whole blood for leukocyte immunophenotype and
- o ADA
- o pSTAT3 (predose [trough] samples only in Phase 1b)
- o CCI
- o CCI
- o CCI
- O See Table 1 and Table 2 for details of PK sampling in the MAD and POC portions
- o Urine pregnancy test will be collected on WOCBP prior to study drug administration
- Spot urine for protein/creatinine ratio
- o Urinalysis
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Full physical examination
- Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours postdose on Day 0)
- 12-lead ECG (prior to PK blood draw)
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, PGA)
- SLICC/ACR damage index
- Study drug administration:
  - Administration of BOS161721 or placebo will take place on-site, and is discussed in Section 7.3
- Injection site reaction assessment performed at 2 hours postdose

Procedures on Day 0 are listed in the Schedule of Assessments (Section 3.4), and details are provided in Section 6.

All patients who are enrolled, randomized, and receive study drug, or undergo study-specific procedures should reconsent with any updated versions of IRB/IEC approved informed consents during study participation as applicable and per institutional guidelines.

# 5.3 Treatment Period/Follow-Up Visits

The following procedures will be performed as indicated in the Schedule of Assessments (Table 1 and Table 2). See Schedule of Assessment tables for allowable windows for each visit.

- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)

• PROs: CCI


Clinical Study Protocol: BOS161721-02


• Urine pregnancy tests will be collected on WOCBP prior to study drug administration

- Injection site reaction assessments will be performed predose
- Direct Coomb's test (if indicated for hemolytic anemia)
- Spot urine for protein to creatinine ratio
- Urinalysis
- CCI
- Plasma CCI
- PGA, BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, and the CLASI will be completed
- SLICC/ACR Damage Index will be completed at Day 180
- C-SSRS
- ECGs prior to PK blood draw
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies, respectively
- Fasting hematology and chemistry assessments
- The CD4+ count and total IgG and IgM levels
- Plasma CC & CC , ADA, and whole blood for leukocyte immunophenotype
- pSTAT3 (predose [trough] samples only Phase 1b)
- nAb will be analyzed by central lab if patient is positive for ADA
- CRP
- CCI

# 5.4 Safety Follow-Up Visits

Safety follow-up visits will take place at Days 210, 240, and 270. These visits will include the following assessments as indicated in the Schedule of Assessments (Table 1 and Table 2):

- PROs: CC
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Injection site reactions
- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Spot urine for protein/creatinine ratio and urinalysis
- Concomitant medication documentation
- BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, and PGA
- Fasting clinical laboratory assessments (hematology and clinical chemistry)
- Direct Coomb's test (if indicated for hemolytic anemia)
- Plasma CC
- · CCI
- 12-lead ECG (prior to PK blood draw)


Clinical Study Protocol: BOS161721-02


- CRP
- ADA
- CCI
- Urine pregnancy test
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC portions, respectively

### 5.5 Premature Discontinuation

While patients are encouraged to complete all study evaluations, they may withdraw from the study at any time and for any reason. Every effort will be made to determine why any patient withdraws from the study prematurely. If the patient is unreachable by telephone, a registered letter, at the minimum, should be sent to the patient requesting him/her to contact the clinic.

All patients who withdraw from the study with an ongoing AE or SAE must be followed until the end of study or until the event is resolved or deemed stable, respectively.

If a patient withdraws prematurely after dosing, an end of treatment (EOT) visit should be performed (Day 180) and a last follow-up visit 90 days after dosing should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 5.4).

Patient participation may be terminated prior to completing the study and the reason recorded as follows:

- AE/SAE
- Protocol deviation
- Lost to follow-up
- Patient withdraws consent at their own request
- Investigator decision
- Decision by sponsor (other than AE/SAE, protocol deviation, or lost to follow-up)

Withdrawn patients may be replaced after discussion between the investigator or designee and sponsor.

### 6 ASSESSMENTS

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances, outside of the control of the investigator, which may make it unfeasible to perform the test. In these cases, the investigator will take all steps necessary to ensure the safety and wellbeing of the patient. When a protocol required test cannot be performed the investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. All protocol violations are entered directly into the eCRFs.


Clinical Study Protocol: BOS161721-02


# 6.1 Medical History, Demographic and Other Baseline Information

The medical history comprises:

- General medical history
- Documentation of SLE diagnosis
- Historical medication therapy for SLE

The following demographic information will be recorded:

- Age
- Ethnic origin (Hispanic/Latino or not Hispanic/not Latino)
- Race (White, American Indian/Alaska Native, Asian, Native Hawaiian or other Pacific Islander, Black/African American)
- Height (without shoes, in cm)
- Body weight, without shoes (kg)
- Body mass index (BMI [kg/m²])

Other baseline characteristics will be recorded as follows:

- Concomitant medication documentation (see Section 4.6)
- Status of child bearing potential and contraception

# **6.2** Safety Assessments

### **6.2.1** Laboratory Assessments

Laboratory tests will be performed at times defined in the Schedule of Assessments (Section 3.4). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

A central laboratory will be used (with the exception of urine pregnancy tests) to ensure accuracy and consistency in test results. Laboratory/analyte results that could unblind the study (ie, biomarker results) will not be reported to investigative sites. Urinalysis will be performed on midstream, clean catch specimens. Some biomarkers listed above will not be drawn at some sites due to geographical logistical challenges. See the laboratory manual for details.

Endpoint analyses will be based on changes from baseline assessments at Days 120 and 210.

Table 3. Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| Hemoglobin | BUN | pН | Spot urine for protein/creatinine ratio |
| Hematocrit | Creatinine | Glucose (qual) | $FSH^b$ |
| RBC count | Glucose (fasting) | Protein (qual) | Urine pregnancy test <sup>c</sup> |
| RDW | Calcium | Blood (qual) | QuantiFERON®-TB Gold In-Tube test |


**Table 3.** Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| MCV | Sodium | Ketones | (QFT-G) <sup>d</sup> |
| MCH | Potassium | Nitrites | Serology <sup>d</sup> (Hepatitis B and C; HIV-1/2 |
| MCHC | Chloride | Leukocyte esterase | combination) |
| Platelet count | Total CO <sub>2</sub> (bicarbonate) | Urobilinogen | Stool sample <sup>e</sup> |
| WBC count | AST, ALT | Urine bilirubin | Serum pregnancy test |
| CD4+ count | Total bilirubin | Microscopy <sup>a</sup> | |
| Total neutrophils | Alkaline phosphatase | | |
| (Abs) | Creatine kinase | | |
| Eosinophils (Abs) | Uric acid | | |
| Monocytes (Abs) | Albumin | | |
| Basophils (Abs) | Total cholesterol | | |
| Lymphocytes (Abs) | (fasting) | | |
| | LDL-C (fasting) | | |
| | HDL-C (fasting) | | |
| | Triglycerides (fasting) | | |
| | Total protein | | |
| | PT/INR | | |
| | Additional Tests <sup>f</sup> | | Immunogenicity, PD and other |
| | (potential Hy's Law) | | Biomarker Tests |
| | AST, ALT (repeat) | | ADA |
| | Total bilirubin (repeat) | | $nAb^g$ |
| | Albumin (repeat) | | pSTAT3 (predose [trough] samples |
| | Alkaline phosphatase | | only in Phase 1b) |
| | (repeat) | | Total IgG & IgM |
| | Direct bilirubin | | Plasma <mark>CCl</mark> |
| | Indirect bilirubin | | Plasma CCI & CCI |
| | GGT | | Whole blood for leukocyte |
| | Prothrombin | | immunophenotype |
| | time/international | | CCI |
| | normalized ratio (repeat) | | CCI |
| | Creatine kinase (repeat) | | CCI |

Abbreviations: Abs = absolute; ADA = anti-drug antibody; ALT = alanine aminotransferase;

CCI ; AST = aspartate aminotransferase; BUN = blood urea nitrogen; C = complement; CD4+ = cluster of differentiation 4; CRP = C-reactive protein; dsDNA = double-stranded deoxyribonucleic acid;; FSH = follicle stimulating hormone; GGT = gamma-glutamyltransferase; HDL-C = high-density lipoprotein cholesterol; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; INR = international normalized ration; IL-21 = interleukin 21; LDL-C = low-density lipoprotein cholesterol; MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = Mean corpuscular volume; nAb = neutralizing antibody; pSTAT3 = phosphorylated signal transducer and activator of transcription 3;

CRP

Direct Coomb's testh

nAb = neutralizing antibody; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; PT = prothrombin time; qual = qualitative; RBC = red blood cell; RDW = RBC distribution width; SAE = serious adverse event; SC = subcutaneous; CC ; TB = tuberculosis.

a. On all urine samples.

c. For WOCBP.


b. At screening only, in women who are amenorrheic for at least 12 consecutive months and under 55 years old.

Clinical Study Protocol: BOS161721-02


**Table 3.** Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|------------|-----------|------------|--------------------|

- d. Screening only.
- e. At screening, and if a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- f. Additional testing for potential Hy's Law cases only (See Section 6.2.2.6.3).
- g. If patient is positive for ADA.
- h. If clinically indicated for hemolytic anemia.

## 6.2.1.1 Pregnancy testing

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, at the last follow up visit day (Day 270) and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures (see Section 5.4) are specified in the Schedule of Assessments (see Section 3.4).

See Section 6.2.2.7.1 for information on reporting of pregnancies as AEs/SAEs during the study.

### **6.2.1.2** Tuberculosis Screening

During the screening period, it must be determined and documented that a patient does not have evidence of active or latent or inadequately treated TB per the exclusion criteria (Section 4.5). The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).

## 6.2.1.2.1 Mycobacterium Tuberculosis Testing Using QuantiFERON Test<sup>40</sup>

QuantiFERON®-TB Gold In-Tube (QFT-G) is an *in vitro* diagnostic test using a peptide cocktail simulating ESAT-6, CFP-10, and TB 7.7 proteins to stimulate cells in heparinized whole blood. Detection of INFγ performed by enzyme-linked immunosorbent assay (ELISA) is used to identify *in vitro* responses to these peptide antigens that are associated with Mycobacterium tuberculosis infection. QFT-G is an indirect test for M. tuberculosis infection (including disease) and is intended for use in conjunction with risk assessment, radiography and other medical and diagnostic evaluations.

Test results will be reported as positive, negative, or indeterminate. A negative QFT-G test result is required to meet the inclusion criterion. In the case of an indeterminate result, repeat tests should be permitted for the purpose of determining eligibility of patients to enroll in this study. If a repeat test is indeterminate again, the patient is a screen failure. The procedure for


Clinical Study Protocol: BOS161721-02


using this test and interpreting the results will be described fully in the laboratory manual, which will be provided to investigators.

#### **6.2.2** Adverse Events

#### 6.2.2.1 Definitions

An AE is defined as any untoward medical occurrence experienced by a study patient, whether or not considered drug related by the principal investigator.

AEs are unfavorable changes in a general condition, subjective or objective signs or symptoms, worsening of pre-existing concomitant disease, and clinically significant abnormality in laboratory parameters observed in a patient in the course of a clinical study.

Non-serious SLE manifestations or abnormal laboratory results related to SLE disease activity would not be recorded as AEs unless they meet the definition for SAEs (Section 6.2.2.5).

## **6.2.2.2** Recording of Adverse Events

AEs should be collected and recorded for each patient from the date of the first dose of study drug until the end of their participation in the study, including the safety follow up period.

AEs may be volunteered spontaneously by the study patient, or discovered by the study staff during physical examinations or by asking an open, nonleading question such as 'How have you been feeling since you were last asked?' All AEs and any required remedial action will be recorded on the Adverse Events eCRF and Safety Adverse Event Form. The details of the AE, date of AE onset, date of AE outcome, and action taken for the AE will be documented together with the principal investigator's assessment of the seriousness of the AE and causal relationship to the study drug and/or the study procedure.

All AEs should be recorded individually, using diagnostic terms where possible. If the diagnosis is not established, individual symptoms may be reported. The AEs will subsequently be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

### **6.2.2.3** Severity of Adverse Events

Each AE will be assessed by the principal investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 criteria. <sup>41</sup> When changes in the severity (grade) of an AE occur more frequently than once a day, the maximum severity for the event should be noted for that day. Any change in severity of signs and symptoms over a number of days will be captured by recording a new AE, with the amended severity grade and the date (and time, if known) of the change.

### **6.2.2.4** Causality of Adverse Events

The principal investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (Table 4) should be selected based on medical judgment, considering the definitions below and all contributing factors.


Clinical Study Protocol: BOS161721-02


### **Table 4.** Causality Definitions

| Related | A clinical event, including laboratory test abnormality, occurs in a plausible time relationship to treatment administration and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (dechallenge <sup>a</sup> ) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge <sup>b</sup> procedure if necessary. |
|---|---|
| Unrelated | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative dechallenge and rechallenge information. Typically explained by extraneous factors (eg, concomitant disease, environmental factors, or other drugs or chemicals). |

- Dechallenge: Upon discontinuation of a drug suspected of causing an AE, the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation (positive dechallenge), or the symptoms continue despite withdrawal of the drug (negative dechallenge). Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia).
- Rechallenge: Upon re-administration of a drug suspected of causing an AE in a specific patient in the past, the AE recurs upon exposure (positive rechallenge), or the AE does not recur (negative rechallenge).

An unexpected adverse drug event is any adverse drug event for which the specificity or severity is not consistent with the current IP.

#### **6.2.2.5** Seriousness of Adverse Events

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life threatening; this means that the patient was at risk of death at the time of the event; it does not mean that the event hypothetically might have caused death if it were more severe
- Requires hospitalization or prolongation in existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly or birth defect
- Is other important medical event (see below)

Important medical events that do not result in death, are not life threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such events are:

- Intensive treatment in an emergency room or at home for allergic bronchospasm
- Blood dyscrasias or convulsions that do not result in inpatient hospitalization
- Development of drug dependency or drug abuse


Clinical Study Protocol: BOS161721-02


Hospitalization for elective surgery or routine clinical procedures that are not the result of AE (eg, elective surgery for a pre-existing condition that has not worsened) need not be considered SAEs. If anything untoward is reported during the procedure, that occurrence must be reported as an AE, either 'serious' or 'nonserious' according to the usual criteria.

Suspected unexpected serious adverse reactions (SUSARs) are AEs that are associated with the use of the drug and are serious and unexpected.

### **6.2.2.6** Adverse Events of Special Interest

AEs of special interest in this study include the following:

- 1. Anaphylaxis and serious allergic reactions
- 2. Grades 2 to 5 injection site reaction, including erythema, pain, and induration (See APPENDIX 6)
- 3. Drug Induced Liver Injury (DILI) assessed following Hy's Law
- 4. Malignancy (not including basal cell carcinoma or squamous cell carcinoma of skin)
- 5. Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, disseminated herpes simplex, disseminated tuberculosis, *Aspergillus* sp., *Candida albicans*, *Coccidioides immitis*, *Cryptococcus neoformans*, *Cytomegalovirus*, *Histoplasma capsulatum*, *Isospora belli*, and *Polyomavirus JC polyomavirus*
- 6. Cryptosporidiasis

### 6.2.2.6.1 Anaphylaxis and Serious Allergic Reactions

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria.<sup>42</sup> In the event of anaphylactic reaction or severe/serious hypersensitivity/allergic reaction, the patient must discontinue IP and emergency resuscitation measures implemented. In case of other mild to moderate hypersensitivity reaction, depending on the severity, the investigator may manage in accordance with the standard-of-care.

Anaphylaxis is highly likely when any one of the following 3 criteria is fulfilled:

- 1. Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (eg, generalized hives, pruritus, or flushing, swollen lips-tongue-uvula) and at least 1 of the following:
  - a. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow [PEF], hypoxemia)
  - b. Reduced blood pressure or associated symptoms of end-organ dysfunction (eg, hypotonia [collapse], syncope, incontinence)
- 2. Two or more of the following that occur rapidly after exposure to a likely allergen for that patient (minutes to several hours):
  - a. Involvement of the skin-mucosal tissue (eg, generalized hives, itch-flush, swollen lips-tongue-uvula)


Clinical Study Protocol: BOS161721-02


b. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)

- c. Reduced blood pressure or associated symptoms (eg, hypotonia [collapse], syncope, incontinence)
- d. Persistent gastrointestinal symptoms (eg, crampy abdominal pain, vomiting)
- 3. Reduced blood pressure after exposure to known allergen for that patient (minutes to several hours):
  - a. Systolic blood pressure of less than 90 mm Hg or greater than 30% decrease from the patient's baseline

### **6.2.2.6.2 Injection Site Reactions**

Injection site reactions are to be captured and reported as AEs. These will include Grades 2 to 5 injection site erythema, pain, and induration (see APPENDIX 6), which are also captured as Adverse Events of Special Interest (See Section 6.2.2.6). The investigator should provide a clear description of the observed or reported AE including location and severity. All concomitant treatments used to treat injection site reactions should be recorded and captured in the eCRF, together with the AE of injection site reactions.

## 6.2.2.6.3 Potential Drug-Induced Liver Injury

Abnormal values in AST and/or ALT levels concurrent with abnormal elevations in total bilirubin level that meet the criteria outlined below in the absence of other causes of liver injury are considered potential cases of DILI, and as potential Hy's Law cases, and should always be considered important medical events. If symptoms compatible with DILI precede knowledge of serum chemical test abnormalities, liver enzyme measurements should be made immediately, regardless of when the next visit or monitoring interval is scheduled. In some cases, symptoms may be an early sign of injury and although typically less sensitive than serum enzyme elevations, they may indicate a need for prompt serum testing. An increase in liver enzymes should be confirmed by a repeated test within 48 to 72 hours following the initial test, prior to reporting of a potential DILI event. Patients will continue to have weekly or biweekly liver enzyme measurements until resolution or levels return to baseline.

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 6.2.2.7.2 for reporting details).

Potential DILI is defined as:

1. ALT or AST elevation  $> 3 \times ULN$ 

AND

2. Total bilirubin > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)

**AND** 


Clinical Study Protocol: BOS161721-02


3. No other immediately apparent possible causes of ALT or AST elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic

The patient should return to the investigational site and be evaluated as soon as possible, include laboratory tests, detailed history, and physical assessment. In addition to repeating measurements of AST and ALT, laboratory tests should include albumin, CK, total bilirubin, direct and indirect bilirubin, GGT, prothrombin time (PT)/International Normalized Ratio (INR), and alkaline phosphatase. A detailed history, including relevant information, such as review of ethanol, acetaminophen, recreational drug and supplement consumption, family history, occupational exposure, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and work exposure, should be collected. Further testing for acute hepatitis A, B, or C infection and liver imaging (eg, biliary tract) may be warranted. All cases confirmed on repeat testing as meeting the laboratory criteria defined above, with no other cause for liver function test (LFT) abnormalities identified at the time should be considered potential Hy's Law cases irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal LFTs. Such potential Hy's Law cases should be reported as SAEs.

Study drug discontinuation is considered if there is marked serum AST or ALT elevation or evidence of functional impairment (as indicated by rising bilirubin or INR, which represent substantial liver injury) that is related to study drug. Discontinuation of treatment should be considered if:

- ALT or AST  $> 8 \times ULN$
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks

Discontinuation of treatment must occur if:

- ALT or AST >3 × ULN and (total bilirubin > 2 × ULN or INR > 1.5)
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%)

### 6.2.2.6.4 Malignancy

The identification of a malignancy event will be made by the study site and communicated to the sponsor or designee. AEs should be reported as serious per the criteria in Section 6.2.2.5.

After the first dose of study drug, when there is a decision to biopsy a potentially malignant tumor, lymph node, or other tissue (with the exception of suspected basal cell/squamous cell), the investigator and/or consultant(s) should contact the sponsor clinicians or designee to discuss the issue and any decisions as soon as possible. Basal cell carcinoma or squamous cell carcinoma of skin is not considered an AE of special interest.


Clinical Study Protocol: BOS161721-02


## 6.2.2.6.5 Specific Infections

Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, disseminated herpes simplex, disseminated tuberculosis, *Aspergillus* sp., *Candida albicans*, *Coccidioides immitis*, *Cryptococcus neoformans*, *Cytomegalovirus*, *Histoplasma capsulatum*, *Isospora belli*, or *Polyomavirus JC polyomavirus* will be recorded as AEs of special interest.

Cryptosporidiosis is also considered an AE of special interest. Patients will be evaluated for cryptosporidium in the stool at screening, and as clinically indicated (eg, watery diarrhea) during the study. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

## **6.2.2.7** Reporting of Adverse Events

AE reporting will be carried out in accordance with applicable local regulations, including regulatory agency and IRB reporting requirements.

Each AE is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

## **6.2.2.7.1** Reporting of Pregnancy

As information is available, a pregnancy diagnosed during the study will be reported within 24 hours to the sponsor via the Pregnancy Notification and Outcome Form, including pregnancy in female patients who received study drug and female partners of male study patients who received study drug. The pregnancy should be followed to term and/or outcome and this outcome should also be reported to the sponsor via the Pregnancy Notification and Outcome Form. Pregnancy itself is not regarded as an AE or SAE unless there is complication.

In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an AE or SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live born, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as serious


Clinical Study Protocol: BOS161721-02


adverse events when the investigator assesses the neonatal death as related or possibly related to exposure to investigational product.

## **6.2.2.7.2** Reporting of Serious Adverse Events

The principal investigator is responsible for providing notification to the sponsor of any SAE via the Safety Adverse Event Form, whether deemed study drug related or not, that a patient experiences during their participation in this study within 24 hours of becoming aware of the event.

If an SAE is fatal or life threatening, notification to the sponsor must be made aware immediately, irrespective of the extent of available AE information. This timeframe also applies to additional new information (follow-up) on previously forwarded SAE reports as well as to the initial and follow-up reporting of exposure during pregnancy and exposure via breastfeeding cases. In the rare event that the investigator does not become aware of the occurrence of an SAE immediately (eg, if an outpatient study patient initially seeks treatment elsewhere), the investigator is to report the event within 24 hours after learning of it and document the time of his/her first awareness of the AE.

The principal investigator will review each SAE and evaluate the intensity and the causal relationship of the event to the study drug. All SAEs will be recorded from the time of first dose of study drug through the safety follow-up period (up to Day 270). SAEs occurring after the final follow-up visit and coming to the attention of the principal investigator must be reported only if there is (in the opinion of the principal investigator) reasonable causal relationship with the study drug.

As a minimum requirement, the initial notification should provide the following information:

- Study number
- Patient number
- Details of the SAE (verbatim details are sufficient for immediate notification)
- Criterion for classification as 'serious'
- Causality assessment (which may be updated in a follow-up report when sufficient information is available to make this classification)

Initial reports of SAEs must be followed later with detailed descriptions, including clear photocopies of other documents as necessary (eg, hospital reports, consultant reports, autopsy reports, etc), with the study patient's personal identifiers removed. All relevant information obtained by the principal investigator through review of these documents will be recorded and submitted to the sponsor within 24 hours of receipt of the information. If a new Safety Adverse Event Form is submitted, then the principal investigator must sign and date the form. The sponsor may also request additional information on the SAE, or clarification of omitted or discrepant information from the initial notification, which the principal investigator or an authorized delegate should submit to the sponsor within 24 hours of the request as possible.


Clinical Study Protocol: BOS161721-02


## **6.2.2.7.3** Reporting of Adverse Events of Special Interest

AEs of special interest will be reported to safety immediately or within 24 hours of the site becoming aware of the event and recorded as such on the Adverse Events eCRF and Safety Adverse Event Form.

Potential DILI will be reported based on specifications mentioned in Section 6.2.2.6.3.

Each AE of special interest is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

## **6.2.2.8** Follow Up of Adverse Events

All AEs will be followed up through the safety follow-up visits. All SAEs experienced by a patient, irrespective of the suspected causality, will be monitored until the event has resolved, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the principal investigator and medical monitor, until there is a satisfactory explanation for the changes observed, or until the patient is lost to follow-up.

See Section 6.2.2.7.1 for details related to follow-up of pregnancy. See Section 6.2.2.6.3 for details related to follow-up of potential DILI. See Section 6.2.2.6.4 for details related to follow-up of malignancy.

## 6.2.3 Vital Signs

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (Section 3.4). Vital signs will be assessed on Day 0 at predose and at Day 0, 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq 5$  minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

### 6.2.4 12-Lead Electrocardiograms

ECG will be assessed as specified in the Schedule of Assessments (Section 3.4). ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

The ECG will include all 12 standard leads and a Lead II rhythm strip on the bottom of the tracing. The ECG will be recorded at a paper speed of 25 mm/second. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QT interval corrected for heart rate using Fridericia's formula (QTcF).


Clinical Study Protocol: BOS161721-02


All ECGs must be evaluated by a qualified physician or qualified designee for the presence of abnormalities and will be captured electronically and retained for future evaluation if required, up to the time of the clinical study report (CSR) completion.

### 6.2.5 Physical Examinations

The full physical examination will be completed at screening and Day 0. It includes an assessment of general appearance and evaluation of head, eyes, ears, nose, mouth, throat, neck, thyroid, lymph nodes, and extremities, and dermatologic, respiratory, cardiovascular, gastrointestinal, musculoskeletal, neurologic, and psychiatric systems.

The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Section 3.4). It includes evaluation of patient complaints and SLE disease-related issues, and will exclude the genitourinary system.

## **6.2.6 C-SSRS**

The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed by Columbia University researchers for the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening.<sup>43</sup>

The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Section 3.4). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

#### **6.2.7** Injection Site Reactions

Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (Section 3.4). Local injection site reactions will be assessed at 2 hours postdose at baseline, and predose for each injection after baseline. Injection site reactions should be managed according to the standard of care. Injection site reactions, Grades 2 to 5, are to be reported as AEs of special interest (see Section 6.2.2.7.3).

#### 6.2.8 Immunogenicity

The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (Section 3.4). Blood samples (4 mL) to provide approximately 1.5 mL of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K<sub>2</sub>EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be


Clinical Study Protocol: BOS161721-02


collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only analyzed by a central lab if the patient had a positive ADA on Day 90.

After the first dose, if a patient tests positive in the validated confirmatory ADA assay, a sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay by a central lab.

## **6.3** Efficacy Assessments

All efficacy assessments will be performed at times defined in the Schedule of Assessments (Section 3.4).

#### **6.3.1 SLEDAI-2K**

The SLEDAI-2K is a validated instrument that measures disease activity in SLE patients at the time of the visit and in the previous 30 days. It is a global index and includes 24 clinical and laboratory variables that are weighted by the type of manifestation, but not by severity. The total score falls between 0 and 105, with higher scores representing increased disease activity. The SLEDAI-2K has been shown to be a valid and reliable disease activity measure in multiple patient groups. A SLEDAI -2K of 6 or more generally represents moderately to severely active disease. 44

#### 6.3.2 BILAG 2004

The BILAG-2004 index is an organ-specific 97-question assessment based on the principle of the doctor's intent to treat. Only clinical features attributable to SLE disease activity are to be recorded and based on the patient's condition in the last 4 weeks compared with the previous 4 weeks. It will be scored as not present (0), improved (1), the same (2), worse (3), or new (4). Disease activity is graded separately for 9 body systems to 5 different grades (A to E) as follows: A ("Active") is very active disease, B ("Beware") is moderate activity, C ("Contentment") is mild stable disease, D ("Discount") is inactive now but previously active, and E ("Excluded") indicates the organ was never involved. A shift from BILAG-2004 Grade A or B to a lower grade indicates a clinically relevant change in disease activity as the BILAG-2004 grades mirror the decision points for treatment interventions.

Only investigators that complete BILAG-2004 training will be allowed to perform the BILAG-2004 assessments. Preferably, the same investigator should evaluate the patient at each BILAG-2004 assessment from screening to study completion. The investigator must maintain documentation with descriptive details supporting the BILAG-2004 scoring (eg, chart, worksheet, clinic notes, and labs) at each visit.

See APPENDIX 5 for detailed specifications.

### 6.3.3 PGA of Disease Activity

The PGA is used to assess investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic


Clinical Study Protocol: BOS161721-02


and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients". PGA worsening is defined as an increase of  $\geq$  30 mm from baseline.

When scoring the PGA, the assessor should always look back at the score from the previous visit.

### 6.3.4 Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response

### **6.3.4.1 SRI-4 Response**

The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. Response based on the SRI-4 is defined by:

1)  $\geq$  4-point reduction in SLEDAI-2K global score, 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B), and 3) no deterioration from baseline in the PGA by  $\geq$  30 mm. The SRI-4 response in patients with moderate to severe SLE is associated with broad improvements in clinical and patient-reported outcomes.<sup>45</sup>

## 6.3.4.2 SRI-5 and SRI-6 Response

Like the SRI-4, the SRI-5 and SRI-6 are composite indices of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. However, the SRI-5 and SRI-6 are computed with a minimal five-point or six-point improvement in SLEDAI-2K being required, respectively. 46

### 6.3.4.3 BICLA Response

The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and PGA. BICLA response is defined as 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (eg, all B [moderate disease] scores falling to C [mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4)  $\leq$  10% deterioration in PGA score and 5) no treatment failure. 44 It is driven primarily by the BILAG, and has been used in Phase 2 and 3 mAb studies. 47

For the endpoints of BICLA response at Days 210, 240, and 270, patient scores will be completed and response determined.

#### 6.3.5 CLASI Response

The CLASI is a comprehensive tool for assessment of disease activity and damage in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity. <sup>48</sup> Response is defined as 50% improvement from baseline in "A" or "B" scores. This assessment will be applied to all patients as all are required to have cutaneous disease activity.

For the secondary efficacy endpoint of CLASI response at Day 210, patient scores on MAD and POC studies will be compared with baseline for 50% improvement.


#### 6.3.6 ACR-28 Joint Count

The ACR-28 joint count will evaluate the number of tender and swollen joints in the shoulder, elbow, wrist, hand, knee joints. Joints of the feet are excluded.

#### 6.4 Other Variables

## 6.4.1 SLICC/ACR Damage Index

The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in patients with SLE regardless of cause, with demonstrated content, face, criterion, and discriminant validity. It will be performed on Days 0 and 180.

### 6.4.2 **PROs**

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the CCI and the CCI and will be assessed as specified in the Schedule of Assessments (Section 3.4).



#### 6.5 Pharmacokinetic Assessments

During the MAD Phase 1b (all sites) and POC Phase 2 (select sites only) parts of the study, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to Table 1 and Table 2.

Plasma concentrations of BOS161721 will be measured using a validated immunoassay. The PK parameters will be calculated from the plasma concentration actual time profiles.

## 6.6 Pharmacodynamic Assessments

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (Section 3.4) for each of the following parameters:

• pSTAT3 (predose [trough] samples only Phase 1b)

• Antibodies: CC

• Plasma complement (CCI)


Clinical Study Protocol: BOS161721-02


- Plasma CCI and CCI
- Whole blood for leukocyte immunophenotype

## 6.7 Pharmacokinetic/Pharmacodynamic Relationship

Evidence of any PK/PD relationships will be evaluated between BOS161721 plasma concentrations and the available PD endpoints and biomarkers.

#### **6.8** Protocol Deviations

Protocol deviations will be documented during the study.

### 7 STUDY DRUG MANAGEMENT

## 7.1 Description

#### 7.1.1 Formulation



Additional information regarding dose preparation will be provided in a separate Pharmacy Manual.

## 7.1.2 Storage

All supplies of BOS161721 or placebo must be stored in accordance with the manufacturer's instructions. BOS161721 or placebo will be stored in a securely locked area, accessible to authorized persons only, until needed for dosing.

Information regarding storage and dose preparation will be provided in a separate Pharmacy Manual.

# 7.2 Packaging and Shipment

Investigational medicinal products will be supplied by Boston Pharmaceuticals, Inc. Investigational medicinal products will be packaged and labeled according to applicable local and regulatory requirements.

### 7.3 Dose and Administration

Details of dosing are provided in Section 3.1.


Clinical Study Protocol: BOS161721-02


Each unit dose will be prepared by a qualified staff member. The vials of investigational product (IP) will appear identical and will have a "blinded" label on the vials that will state mg or placebo. When the site goes into the IWRS to request the patient kit(s), the IWRS will assign the appropriate number of kits (regardless of assignment to placebo or active treatment) per the dose (ie, CC).

If a patient is randomized to the placebo arm, they will receive the matching number of kits.

The designated staff member (or designee under the direction of the designated staff member) will dispense BOS161721 or placebo for each patient according to the protocol, randomization list, and Pharmacy Manual, if applicable.

After receiving sponsor approval in writing, the investigational site is responsible for returning all unused or partially used BOS161721 or placebo to the sponsor or designated third party or for preparing BOS161721 or placebo for destruction via incineration.

Further details are found in a separate Pharmacy Manual.

## 7.4 Accountability

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Products returned to the pharmacy will be stored under the same conditions as products not yet dispensed. The returned products should be marked as 'returned' and kept separate from the products not yet dispensed.

All dispensing and accountability records will be available for sponsor review after database lock procedures are completed. During safety monitoring, the drug accountability log will be reconciled with the products stored in the pharmacy.

## 7.5 Prohibited Concomitant Therapy

Prohibited concomitant medications are discussed in Section 4.6 and APPENDIX 4 and will be listed as protocol violations if taken when not permitted.

# 7.6 Compliance

Dosing will be performed by trained, qualified personnel designated by the principal investigator. The date and time of dosing will be documented on each dosing day. Comments will be recorded if there are any deviations from the planned dosing procedures.

### 8 STATISTICS

The following analyses are planned:

• An IA will be performed during the last cohort of the MAD portion to determine dose selection for the POC part of the study.


• An additional analysis may be performed for the MAD portion of the study when all MAD patients have completed the safety follow-up or withdrawn from the study, and prior to final analysis. Data from the POC part of the study will be excluded from this additional analysis.

- The final analysis will be performed when all patients have completed the POC safety follow-up or withdrawn from the study.
- Safety analyses will be performed for DMC reviews throughout the study to evaluate dose escalation decisions and accumulating safety data. The frequency and details of the content and format of the safety review meetings will be described in the SAP and/or DMC charter.

All statistical analyses will be performed using Statistical Analysis Software (SAS®) Version 9 or higher.

The following standards will be applied for the analysis unless otherwise specified. Data will be summarized descriptively by treatment and overall for each study portion. For the MAD part of the study, BOS161721 will be summarized overall and by each dose level, and placebo patients from each cohort will be combined. Select parameters may be summarized using patients from both study parts. Statistical testing will be performed on data from the Phase 2 portion only.

Continuous data will be summarized using number, mean, standard deviation (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, median, and maximum. Categorical data will be summarized by treatment group using frequency tables (number and percentage). Time to event data will be summarized using counts, medians, 25<sup>th</sup> and 75<sup>th</sup> percentiles, and standard error. All data will be listed for all patients.

Statistical inference will be based on a 2-tailed test with an overall 0.10 level of significance, unless stated otherwise.

The effects of noncompliance, background therapy use, treatment discontinuations, premature withdrawal from study and covariates will be assessed to determine the impact on the general applicability of results from this study. Exploratory analyses of the data will be conducted as deemed appropriate. Any deviations from the planned analyses will be described and justified in the final integrated CSR.

Protocol deviations and prohibited medications that define medication failures will be fully assigned and documented before database lock and unblinding.

Further details of the analysis, including the handling of missing data, transformations and other data handling procedures will be provided in the SAP.

## 8.1 Sample Size

Sample size in the Phase 1b part of the study is based on operational consideration.

The sample size in the Phase 2 portion is based on the primary endpoint, SRI-4 Response at Day 210. Approximately 156 additional patients will be randomized in a 2:1 ratio to BOS161721 versus placebo to achieve 132 evaluable patients in the FAS. This assumes


Clinical Study Protocol: BOS161721-02


24 patients will drop prior to having received treatment and an evaluable post-baseline efficacy measure. Enrollment and randomization will be monitored in a blinded fashion and increased if needed to ensure at least 132 patients are randomized into the FAS.

A total of 132 patients randomized provides more than 80% power to detect a treatment difference of 25% in SRI-4 response rates at Day 210, based on a targeted 2-sided significance level of 10% and using a 2-sided Pearson's chi-squared test. This assumes of a response rate of 65% for BOS161721 and 40% for placebo, where missing data at Day 210 is carried forward from most recent non-missing result and patients are treated as a non-responder if a prohibited medication defined as a medication failure occurs.

#### **8.2** Statistical Methods

### 8.2.1 Analysis Populations

The primary efficacy analysis will be based on the FAS, defined as all patients who receive at least 1 dose of study treatment and at have least 1 evaluable post-baseline efficacy evaluation. FAS analyses will be conducted on the basis of the randomized treatment.

A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be identified based on blinded data prior to study unblinding. PP analyses will be conducted on the basis of the randomized treatment.

Safety analyses will be based on the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. Safety analyses will be conducted on the basis of actual treatment received.

Pharmacokinetic analysis will be conducted on the PK analysis set, defined as the FAS with sufficient concentration data for the calculation of PK parameters.

### 8.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized using all randomized patients.

### 8.2.3 Primary Efficacy Endpoint(s)

The proportion of patients who achieve a SRI-4 response at Day 210 will be assessed via Pearson's chi-squared analysis. The primary efficacy endpoint will be analyzed using the FAS and if needed repeated in the PP analysis set. Missing values will be addressed by employing a last observation carried forward (LOCF) analysis. Other imputation methods may be employed as a sensitivity analysis and will be described in the SAP. Additional analyses exploring impact of baseline factors such as baseline disease severity, race, and other characteristics may be performed.

Patients that received prohibited medications or unallowable CS usage as described in Section 4.6 will be considered "medication failures" and will be treated as non-responders for the


Clinical Study Protocol: BOS161721-02


primary efficacy analysis. The determination of medication failures will be reviewed using blinded data and finalized prior to unblinding.

The superiority of BOS161721 relative to placebo will be evaluated. If the proportion of SRI-4 responders for the selected POC dose in BOS161721 arm is higher than that of the placebo arm, then BOS161721 will be considered superior to placebo if the 2-sided p-value is less than 0.10. Secondary and exploratory endpoints for this POC portion will be evaluated based on the same statistical hypothesis.

### 8.2.4 Secondary Efficacy Endpoint(s)

Binary efficacy endpoints will be assessed via Pearson's chi-squared analysis. Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) and treatment will be compared using the F-test. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test. The secondary efficacy endpoints will be analyzed on the FAS and if needed repeated in the PP analysis set. Details including handling of missing data and "medication failures" will be available in the SAP.

#### 8.2.5 Analysis of Safety

## 8.2.5.1 Safety Analysis

Safety analyses will be performed on the SS. AE data will be coded to system organ class and preferred term using MedDRA. The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term, will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be coded using the WHO Drug dictionary. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters will be summarized at each individual visit.

#### 8.2.6 Pharmacokinetic and Pharmacodynamic Data

### 8.2.6.1 Analysis of Pharmacokinetic Data

PK parameters will be calculated from concentration data collected during the MAD Phase 1b portion of the study using non-compartmental analysis and include the following:

• C<sub>max</sub>, T<sub>max</sub>, AUC, t<sub>1/2</sub>, CL, V<sub>d</sub>

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:

• A listing of all plasma BOS161721 concentrations by patient at actual times post dose;


Clinical Study Protocol: BOS161721-02


• A descriptive summary of plasma BOS161721 concentrations. Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.

## 8.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Exploratory analyses examining the relationship between PD parameters and PK concentration and PK parameters will be performed.

## 8.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints.

## 8.3 Interim Analysis and Power

One IA is planned for this study and will be conducted at the time of the POC decision for dose selection.

Since there is no IA during the POC part of the study, there is no impact on the type 1 error.

## 9 ETHICS AND RESPONSIBILITIES

#### 9.1 Good Clinical Practice

The procedures set out in this protocol are designed to ensure that the sponsor and the principal investigator abide by the principles of the International Council for Harmonisation (ICH) guidelines on GCP and the Declaration of Helsinki (Version 2013). The clinical study also will be carried out in the keeping with national and local legal requirements (in accordance with US IND regulations [21 CFR 56]).

### 9.2 **DMC**

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for BOS161721. The recommendations made by the DMC (ie, dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.


The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) suggest dose for POC portion of the study as described in Section 3.1.1.3.

The DMC considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

The DMC will have access to unblinded treatment information during the clinical trial. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of BOS161721 treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.

#### 9.3 Institutional Review Board/Independent Ethics Committee

Independent Ethics Committees/IRB must meet the guidelines set out by the U.S. Food and Drug Administration (FDA) and conform to local laws and customs where appropriate. Written IRB/IEC approval for the protocol and the signed ICF must be obtained and transmitted to Boston Pharmaceuticals or representative before the study can be initiated. The IRB/IEC must be informed of and approve all protocol amendments. The investigator will ensure that this study is conducted in full conformance with all applicable local and regional laws and regulations. The complete text of the World Medical Association Declaration of Helsinki is given in APPENDIX 2.

#### 9.4 Informed Consent

Before each patient undergoes any protocol required assessments or procedure, the written informed consent will be obtained according to the regulatory and legal requirements of the participating country. As part of this procedure, the principal investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study patient should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The principal investigator or designee will provide the sponsor with a copy of the IRB-approved ICF prior to the start of the study.

The informed consent document must be signed and dated; 1 copy will be handed to the patient and the principal investigator will retain a copy as part of the clinical study records. The principal investigator will not undertake any investigation specifically required for the clinical


Clinical Study Protocol: BOS161721-02


study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented.

If the informed consent document is revised, it must be reviewed and approved by the responsible IRB/IEC. Patients currently enrolled may need to sign this revision (based on IRB/IEC requirements) and all future patients enrolled in the clinical study will be required to sign this revised ICF.

#### 9.5 Records Management

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes. The principal investigator or designee will cooperate with the sponsor's representative(s) for the periodic review of study documents to ensure the accuracy and completeness of the data capture system at each scheduled monitoring visit.

Electronic consistency checks and manual review will be used to identify any errors or inconsistencies in the data. This information will be provided to the respective study sites by means of electronic or manual queries.

The principal investigator or designee will prepare and maintain adequate and accurate study documents (medical records, ECGs, AE and concomitant medication reporting, raw data collection forms, etc.) designed to record all observations and other pertinent data for each patient receiving BOS161721 or placebo.

The principal investigator will allow sponsor representatives, contract designees, authorized regulatory authority inspectors, and the IRB to have direct access to all documents pertaining to the study.

Electronic case report forms are required and should be completed for each randomized patient. It is the principal investigator's responsibility to ensure the accuracy, completeness, legibility, and timeliness of the data reported on the patients' eCRF. Electronic case report forms should be completed in a timely fashion to support the study timelines. Source documentation supporting the eCRF data should indicate the patient's participation in the study and should document the dates and details of study procedures, AEs, and patient status. The principal investigator or designated representative should complete and the principal investigator should verify the source documents as the information is collected. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the Sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes.


Clinical Study Protocol: BOS161721-02


#### 9.6 Source Documentation

The documents that will form the source data for the clinical study (eg, patient charts, laboratory reports) must be defined and documented in the in-house study master file prior to the start of the study. Data on the eCRFs which will be checked against source data during monitoring visits must also be defined and documented in the in-house study master file including the percentage of each of the source data to be verified and the percentage of patients' eCRFs to be monitored.

## 9.7 Study Files and Record Retention

According to ICH guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of BOS161721. However, these documents should be retained for a longer period if required by the applicable legal requirements.

#### 10 AUDITING AND MONITORING

Throughout the course of the study, the study monitor will make frequent contacts with the investigator. This will include telephone calls and on-site visits. The study will be routinely monitored to ensure compliance with the study protocol and the overall quality of data collected. During the on-site visits, the eCRFs will be reviewed for completeness and adherence to the protocol. As part of the data audit, source documents will be made available for review by the study monitor. The study monitor may periodically request review of the investigator study file to assure the completeness of documentation in all respects of clinical study conduct. The study monitor will verify that each patient has proper consent documentation from the patient and/or patient's authorized representative for study procedures and for the release of medical records to the sponsor, FDA, other regulatory authorities, and the IRB. The study monitor will also verify that assent was obtained for patients not capable of providing informed consent or that documentation is provided by the investigator explaining why the patient was unable to provide assent. The investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the investigator will permit inspection of the study files by authorized representatives of the regulatory agencies. On completion of the study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

Throughout the course of the study, the medical monitor will determine eligibility of all screened patients, will address any medical issues that might arise, clarify medical questions, review patient safety data (eg, AE/SAE, laboratory, and ECG), and partner with the study team in the overall study management. The study medical monitoring plan will document additional details of the study medical oversight and monitoring.

#### 11 AMENDMENTS

Protocol modifications, except those intended to reduce immediate risk to study patients, may be made only by Boston Pharmaceuticals. A protocol change intended to eliminate an apparent


Clinical Study Protocol: BOS161721-02


immediate hazard to patients may be implemented immediately, provided the IRB/IEC is notified within 5 days.

Any permanent change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB/IEC and the investigator must await approval before implementing the changes. Boston Pharmaceuticals will submit protocol amendments to the appropriate regulatory authorities for approval.

If in the judgment of the IRB/IEC, the investigator, and/or Boston Pharmaceuticals, the amendment to the protocol substantially changes the study design and/or increases the potential risk to the patient and/or has an impact on the patient's involvement as a study participant, the currently approved written ICF will require similar modification. In such cases, informed consent will be renewed for patients enrolled in the study before continued participation.

#### 12 STUDY REPORT AND PUBLICATIONS

Boston Pharmaceuticals is responsible for preparing and providing the appropriate regulatory authorities with clinical study reports according to the applicable regulatory requirements.

By signing the protocol, the principal investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the principal investigator's name, address, qualifications, and extent of involvement.

The principal investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted and obtained approval from the sponsor in advance.

#### 13 STUDY DISCONTINUATION

Both Boston Pharmaceuticals and the principal investigator reserve the right to terminate the study at the investigator's site at any time. Should this be necessary, Boston Pharmaceuticals or a specified designee will inform the appropriate regulatory authorities of the termination of the study and the reasons for its termination, and the principal investigator will inform the IRB/IEC of the same. In terminating the study Boston Pharmaceuticals and the principal investigator will assure that adequate consideration is given to the protection of the patients' interests.

#### 14 CONFIDENTIALITY

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from Boston Pharmaceuticals, except to the extent necessary to obtain informed consent from patients who wish to participate in the trial or to comply with regulatory requirements. However, authorized regulatory officials, IRB/IEC personnel, Boston Pharmaceuticals, and its authorized representatives are allowed full access to the records.

Identification of patients and eCRFs shall be by initials, birthdate, or patient number. Documents that identify the patient (eg, the signed informed consent document) must be


Clinical Study Protocol: BOS161721-02


maintained in confidence by the principal investigator. If required, the patient's full name may be made known to an authorized regulatory agency or other authorized official.


#### 15 REFERENCES

1 Urowitz MB, Gladman DD. How to improve morbidity and mortality in systemic lupus erythematosus. Rheumatology 2000;39:238-44.

- 2 Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, et al. Morbidity and Mortality in Systemic Lupus Erythematosus During a 10-Year Period. Medicine 2003;82(5):299-308.
- 3 Pons-Estel GJ, Alarcón GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010;39(4):257. Epub 2009 Jan 10.
- 4 Kanta H, Mohan C. Three Checkpoints in lupus development: central tolerance in adaptive immunity, peripheral amplification by innate immunity, and end-organ inflammation. Genes and Immunity 2009;10:390-6.
- 5 Dall'Aqua WF, Kiener PA, Wu H. Properties of Human IgG1s Engineered for Enhanced Binding to the Neonatal Fc Receptor (FcRn). J Biol Chem. 2006 Aug 18, 281(33):23514-24.
- 6 Spolski R, Leonard WJ. The Yin and Yang of interleukin-21 in allergy, autoimmunity and cancer. Curr Opin Immunol. 2008a;20:295-301.
- 7 Asao H, Okuyama C, Kumaki S, Ishii N, Tsuchiya S, Foster D, et al. Cutting edge: the common gamma-chain is an indispensable subunit of the IL-21 receptor complex. J Immunol. 2001;167:1-5.
- 8 Habib T, Senadheera S, Weinberg K, Kaushansky K. The common gamma chain (gamma c) is a required signaling component of the IL-21 receptor and supports IL-21-induced cell proliferation via JAK3. Biochemistry. 2002;41:8725-31.
- 9 Spolski R, Leonard WJ. Interleukin-21: basic biology and implications for cancer and autoimmunity. Annu Rev Immunol. 2008b;26:57-79.
- 10 Puga I, Cols M, Barra CM, He B, Cassis L, Gentile M, et al. B-cell-helper neutrophils stimulate the diversification and production of immunoglobulin in the marginal zone of the spleen. Nat Immunol. 2011;13(2):170-80.
- 11 Costanzo A, Chimenti MS, Botti E, Caruso R, Sarra M, Monteleone G. IL-21 in the pathogenesis and treatment of skin diseases. J Dermatol Sci. 2010;60(2):61-6.
- 12 Avery DT, Bryant VL, Ma CS, de Waal Malefy R, Tangye SG. IL-21-induced isotype switching to IgG and IgA by human naive B cells is differentially regulated by IL-4. J Immunol. 2008;181:1767-79.
- 13 Rasmussen TK, Andersen T, Bak, RO, Yiu G, Sorensen CM, Stengaard-Pedersen K, et al. Overexpression of microRNA-155 increases IL-21 mediated STAT3 signaling and IL-21 production in systemic lupus erythematosus. Arthritis Research & Therapy 2015;17(154)


14 Ettinger R, Kuchen S, Lipsky PE. The role of IL-21 in regulating B-cell function in health and disease. Immunol Rev. 2008;223:60-86.

- 15 Caprioli F, Sarra M, Caruso R, Stolfi C, Fina D, Sica G, et al. Autocrine regulation of IL-21 production in human T lymphocytes. J Immunol. 2008;180(3):1800-7.
- 16 Yang L, Anderson DE, Baecher-Allan C, Hastings WD, Bettelli E, Oukka M, et al. IL-21 and TGF-beta are required for differentiation of human T(H)17 cells. Nature. 2008;454(7202):350-2.
- 17 Tangye SG, Ma CS, Brink R, Deenick EK. The good, the bad and the ugly TFH cells in human health and disease. Nat Rev Immunol. 2013;13(6):412-26.
- 18 Fantini MC, Rizzo A, Fina D, Caruso R, Becker C, Neurath MF, et al. IL-21 regulates experimental colitis by modulating the balance between Treg and Th17 cells. Eur J Immunol. 2007;37(11):3155-63.
- 19 Peluso I, Fantini MC, Fina D, Caruso R, Boirivant M, MacDonald TT, et al. IL-21 counteracts the regulatory T-cell-mediated suppression of human CD4+ T lymphocytes. J Immunol. 2007;178(2):732-9.
- 20 Hippen KL, Bucher C, Schirm DK, Bearl AM, Brender T, Mink KA, et al. Blocking IL-21 signaling ameliorates xenogeneic GVHD induced by human lymphocytes. Blood. 2012;119(2):619-28.
- 21 Davis ID, Skrumsager BK, Cebon J, Nicholaou T, Barlow JW, Moller NP, et al. An open-label, two-arm, phase I trial of recombinant human interleukin-21 in patients with metastatic melanoma. Clin Cancer Res. 2007;13:3630-6.
- 22 Frederiksen KS, Lundsgaard D, Freeman JA, Hughes SD, Holm TL, Skrumsager BK, et al. IL-21 induces in vivo immune activation of NK cells and CD8(+) T-cells in patients with metastatic melanoma and renal cell carcinoma. Cancer Immunol Immunother. 2008;57(10):1439-49.
- 23 Karrich JJ, Jachimowski LC, Nagasawa M, Kamp A, Balzarolo M, Wolkers MC, et al. IL-21- stimulated human plasmacytoid dendritic cells secrete granzyme B, which impairs their capacity to induce T-cell proliferation. Blood. 2013;121(16):3103-11.
- 24 Lindner S, Dahlke K, Sontheimer K, Hagn M, Kaltenmeier C, Barth TF, et al. Interleukin-21-induced granzyme B-expressing B-cells infiltrate tumors and regulate T-cells. Cancer Res. 2013;73(8):2468-79.
- 25 Monteleone G, Caruso R, Fina D, Peluso I, Gioia V, Stolfi C, et al. Control of matrix metalloproteinase production in human intestinal fibroblasts by interleukin 21. Gut. 2006;55(12):1774-80.
- 26 Nakou M, Papadimitraki ED, Fanouriakis A, Bertsias GK, Choulaki C, Goulidaki N, et al. Interleukin-21 is increased in active systemic lupus erythematosus patients and contributes to the generation of plasma B-cells. Clin Exp Rheumatol. 2013;31(2):172-9.


27 Li Q, Liu Z, Dang E, Jin L, He Z, Yang L, et al. Follicular helper T-cells (Tfh) and IL-21 involvement in the pathogenesis of bullous pemphigoid. PLoS One. 2013;8(7):e68145.

- 28 Liu R, Wu Q, Su D, Che N, Chen H, Geng L, et al. A regulatory effect of IL-21 on T follicular helper-like cell and B-cell in rheumatoid arthritis. Arthritis Res Ther. 2012;14(6):R255.
- 29 Kang KY, Kim HO, Kwok SK, Ju JH, Park KS, Sun DI, et al. Impact of interleukin-21 in the pathogenesis of primary Sjögren's syndrome: increased serum levels of interleukin-21 and its expression in the labial salivary glands. Arthritis Res Ther. 2011;13(5):R179.
- 30 Terrier B, Geri G, Chaara W, Allenbach Y, Rosenzwajg M, Costedoat-Chalumeau N, et al. Interleukin-21 modulates Th1 and Th17 responses in gianT-cell arteritis. Arthritis Rheum. 2012a;64(6):2001-11.
- 31 Terrier B, Costedoat-Chalumeau N, Garrido M, Geri G, Rosenzwajg M, Musset L, et al. Interleukin 21 correlates with T-cell and B-cell subset alterations in systemic lupus erythematosus. J Rheumatol. 2012b;39(9):1819-28.
- 32 International Conference on Harmonisation. Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals S6 (R1). 2011.
- 33 Wang W, Wang EQ, Balthasar JP. Monoclonal Antibody Pharmacokinetics and Pharmacodynamics. Clin Pharm & Ther 2008; 84(5):548-58.
- 34 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 35 Elsaesser H, Sauer K, Brooks DG. IL-21 is required to control chronic viral infection. Science. 2009;324(5934):1569-72
- 36 Kotlarz D, Zietara N, Uzel G, Weidemann T, Braun CJ, Diestelhorst J, et al. Loss-of-function mutations in the IL-21 receptor gene cause a primary immunodeficiency syndrome. J Exp Med. 2013;210(3):433-43.
- 37 Hunter PR, Nichols G. Epidemiology and clinical features of Cryptosporidium infection in immunocompromised patients. Clinical microbiology reviews. 2002;15(1):145-54.
- 38 Desjardins M, Mazer BD. B-cell memory and primary immune deficiencies: interleukin-21 related defects. Curr Opin Allergy Clin Immunol. 2013;13(6):639-45.
- 39 Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. *Nephron*. 1976;16(1):31-41.


40 Guidelines for Using the QuantiFERON®-TB Gold Test for Detecting Mycobacterium tuberculosis Infection, US: http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5415a4.htm.

- 41 NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, available at https://evs.nci.nih.gov/ftp1/CTCAE/About.html.
- 42 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 43 Posner K, Melvin G a, Stanley B, Oquendo M a, Gould M. Factors in the assessment of suicidality in youth. *CNS Spectr*. 2007;12(2):156-162.
- 44 Castrejon I, Tani C, Jolly M, Huang A, Mosca M. Indices to assess patients with systemic lupus erythematosus in clinical trials, long-term observational studies, and clinical care. Clin Exp Rheumatol 2014; 32(85):S85-95.
- 45 Furie R, Wang L, Drappa J, Illei G. Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] Response Is Associated with Global Benefit in Patients with Moderate to Severe SLE [abstract]. *Arthritis Rheumatol*. 2016; 68 (suppl 10).
- 46 Thanou A, Chakravarty E, James JA, Merrill JT. Which outcome measures in SLE clinical trials best reflect medical judgment? Lupus Science & Medicine 2014;1:e000005. doi:10.1136/lupus-2013-000005.
- 47 Wallace DJ, Kalunian K, Petri MA, Strand V, Houssiau FA, Pike M, et al. Efficacy and safety of epratuzumab in patients with moderate/severe active systemic lupus erythematosus: results from EMBLEM, a phase IIb, randomised, double-blind, placebo-controlled, multicentre study. *Ann Rheum Dis* 2014;73:183-90.
- 48 Albrecht J, Taylor L, Berlin JA, Dulay S, Ang G, Fakharzadeh S. The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index): An Outcome Instrument for Cutaneous Lupus Erythematosus. J Invest Derm. 2005;125(5):889-94.
- 49 Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is Valid, and Renal and Pulmonary Organ Scores are Predictors of Sever Outcome in Patients with Systemic Lupus Erythematosus. Br J Rheumatol. 1996;35:248-54.

50 **CC** 


# 16 APPENDICES

# APPENDIX 1 NAMES OF STUDY PERSONNEL



Central Laboratory: PPD

PPD


#### APPENDIX 2 DECLARATION OF HELSINKI

## WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI

Ethical Principles
For
Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly
Helsinki, Finland, June 1964
and amended by the
29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
and the

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### A. INTRODUCTION

The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.

It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.

The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my subject will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the subject's interest when providing medical care which might have the effect of weakening the physical and mental condition of the subject."

Medical progress is based on research, which ultimately must rest in part on experimentation involving human subjects.

In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.

The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic, and therapeutic procedures and the understanding of the etiology and pathogenesis of disease. Even the best-proven prophylactic, diagnostic, and therapeutic methods must continuously be challenged through research for their effectiveness, efficiency, accessibility, and quality.


Clinical Study Protocol: BOS161721-02


In current medical practice and in medical research, most prophylactic, diagnostic, and therapeutic procedures involve risks and burdens.

Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.

Research investigators should be aware of the ethical, legal, and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal, or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### B. BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.

Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.

Appropriate caution must be exercised in the conduct of research, which may affect the environment, and the welfare of animals used for research must be respected.

The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any SAEs. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.

The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles enunciated in this Declaration.

Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a subject of the research, even though the subject has given consent.

Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the


subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.

Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.

Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.

Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.

The subjects must be volunteers and informed participants in the research project.

The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the subject's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.

In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.

When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.

For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the investigator must obtain informed consent from the legally authorized representative in accordance with applicable law. These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.

When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the investigator must obtain that assent in addition to the consent of the legally authorized representative.

Research on individuals from whom it is not possible to obtain consent, including proxy or advance consent, should be done only if the physical/mental condition that prevents obtaining


Clinical Study Protocol: BOS161721-02


informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.

Both authors and publishers have ethical obligations. In publication of the results of research, the investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic, or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the subjects who are research subjects.

The benefits, risks, burdens, and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic, or therapeutic method exists.

At the conclusion of the study, every subject entered into the study should be assured of access to the best-proven prophylactic, diagnostic, and therapeutic methods identified by the study.

The physician should fully inform the subject which aspects of the care are related to the research. The refusal of a subject to participate in a study must never interfere with the subject-physician relationship.

In the treatment of a subject, where proven prophylactic, diagnostic, and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the subject, must be free to use unproven or new prophylactic, diagnostic, and therapeutic measures, if in the physician's judgment it offers hope of saving life, re-establishing health, or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases, new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.


# APPENDIX 3 COMMONLY USED CORTICOSTEROID EQUIVALENTS

| Medication | Prednisone Dose Equivalence |
|--------------------|-----------------------------|
| Prednisone | 1 mg |
| Cortisone | 5 mg |
| Hydrocortisone | 4 mg |
| Prednisolone | 1 mg |
| Methylprednisolone | 0.8 mg |
| Triamcinolone | 0.8 mg |
| Budesonide | 0.25 mg |
| Dexamethasone | 0.16 mg |
| Bethamethasone | 0.16 mg |


# APPENDIX 4 MEDICATION WASHOUT PERIODS

## WASHOUT TIMES OF MEDICATIONS BASED ON 5 HALF-LIVES

| Medication | Discontinuing Prior to Signing Consent |
|---|---|
| Abatacept (CTLA4Ig) | 24 weeks |
| Alefacept | 12 weeks |
| AMG 623 (blisibimod) | 24 weeks |
| Anifrolumab | 12 weeks |
| Atacicept (TACI-Ig) | 12 weeks |
| Belimumab | 24 weeks |
| Cyclophosphamide | 24 weeks |
| Cyclosporine (except for CSA eye drops) | 4 weeks for oral and 8 weeks for topical |
| Danazol | 4 weeks |
| Dapsone | 4 weeks |
| Eculizumab | 12 weeks |
| Efalizumab | 12 weeks |
| Epratuzumab | 24 weeks |
| Intravenous globulin | 4 weeks |
| Leflunomide | 8 weeks (4 weeks for washout with |
| | cholestyramine) |
| Lenalidomide with cholestiramine | 8 weeks |
| Lupuzor | 12 weeks |
| Memantine | 4 weeks |
| Natalizumab | 24 weeks |
| Ocrelizumab | 48 weeks (or 24 weeks with recovery of B cell) |
| Pimecrolimus | 4 weeks |
| Plasmapheresis | 24 weeks |
| Retinoids (oral or topical) | 4 weeks |
| Rituximab | 48 weeks (or 24 weeks with recovery of B cell) |
| Sirolimus | 4 weeks |
| Tacrolimus | 4 weeks |
| Thalidomide | 8 weeks |
| Tocilizumab | 12 weeks |


# APPENDIX 5 BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA)




Clinical Study Protocol: BOS161721-02


# APPENDIX 6 INJECTION SITE REACTION GRADING SCALE

| Adverse event Injection site reaction | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade<br>5 |
|---|---|---|---|---|---|
| Definition: A disorder<br>characterized by an<br>intense adverse reaction<br>(usually immunologic)<br>developing at the site of<br>an injection | Tenderness with<br>or without<br>associated<br>symptoms (eg,<br>warmth,<br>erythema,<br>itching) | Pain;<br>Lipodystrophy;<br>Edema;<br>phlebitis | Ulceration or<br>necrosis;<br>Severe tissue<br>damage;<br>Operative<br>intervention<br>indicated | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>indicated | Death |
| Pain | Mild pain | Moderate pain;<br>limiting<br>instrumental ADL | Severe pain;<br>limiting self-<br>care ADL | - | - |
| Rash maculopapular/Erythema /Induration | Macules/papules<br>covering <10%<br>BSA with or<br>without | Macules/papules<br>covering 10% -<br>30% BSA with or<br>without symptoms | Macules/papul<br>es covering<br>> 30% BSA<br>with or | - | - |
| Definition: A disorder<br>characterized by the<br>presence of macules<br>(flat) and papules<br>(elevated). Also known<br>as morbillform rash, it is | symptoms (eg,<br>pruritus, burning,<br>tightness)<br>Erythema<br>covering <10%<br>BSA with or | (eg, pruritus,<br>burning, tightness);<br>limiting<br>instrumental ADL;<br>Erythema 30%<br>BSA with or | without<br>associated<br>symptoms;<br>limiting<br>self-care ADL | | |
| one of the most common<br>cutaneous adverse<br>events, frequently<br>affecting the upper trunk,<br>spreading centripetally,<br>and associated with | without<br>symptoms (eg,<br>pruritus, burning,<br>tightness) | without symptoms<br>(eg, pruritus,<br>burning, tightness);<br>limiting<br>instrumental ADL | Erythema<br>covering<br>> 30% BSA<br>with or<br>without<br>associated | | |
| pruritus. | | | symptoms;<br>limiting<br>self-careADL | | |

ADL = active daily living


Endpoints, Phase 2

Proof of Concept,


# APPENDIX 7 PROTOCOL SUMMARY OF CHANGES

The protocol summary of changes was moved to the end of the protocol for easier readability.

Significant changes are described in the table below. Changed text is displayed for the first major occurrence only. Deleted text is presented in strikethrough format, and added text is presented in bold format.

| Section | Description of Changes | Rationale |
|---|---|---|
| Global | Replace: | Administrative |
| | Protocol Date and Version: 27 July 2018; V4.0 | |
| | With: | |
| Global | Change: | Administrative |
| | Changed Version number from V4.0 (Amendment 3) to V5.0 (Amendment 4) and Version date from 27 July 2018 to 23 January 2019. | |
| Global | Made administrative and editorial (formatting, typographical, and grammatical) updates. | Administrative |
| PROTOCOL SUMMARY, Objectives and Endpoints, MAD Phase 1b, Secondary Objectives Section 2.1, Study Objectives and Endpoints, Phase 1b Multiple Ascending Dose, Secondary Objectives | <ul> <li>Replace: <ul> <li>To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PD effects in patients with mild to moderate SLE.</li> </ul> </li> <li>With: <ul> <li>To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PD effects in patients with moderately to severely active SLE.</li> </ul> </li> </ul> | Error in the previous protocol; text updated to "moderately to severely active." |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints, POC<br>Phase 2, Safety<br>Objectives<br>Section 2.2, Study<br>Objectives and | Replace: • To assess safety and tolerability of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment With: | Error in the previous protocol; text updated to reflect the POC study and not the 3 doses used in the MAD Phase 1b study. |


the chosen dose administered SC in adult patients with

To assess safety and tolerability of repeat doses of BOS161721 at

moderately to severely active SLE on limited background standard


# Section

#### **Description of Changes**

of care treatment

#### Rationale

Safety Objectives

PROTOCOL

#### Replace:

SUMMARY, Objectives and Endpoints, POC

Phase 2, Exploratory Objectives

Section 2.2, Study Objectives and Endpoints, Phase 2 Proof of Concept, Exploratory



With:

Objectives **PROTOCOL** SUMMARY, Study

Design, Paragraph 5

#### Replace:

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 60. Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits. Tapering may occur after randomization except within 60 days of the primary (Day 210) and secondary (Day 120) endpoint assessments. Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant.

Protocol clarification; text was reworded to better explain the importance of tapering when allowed and to reiterate when it is not.

#### With:

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 60. Tapering of steroids during the course of the study will be highly encouraged and should be evaluated at the protocol permitted visits (Day 0 through Day 60 and Day 120 through Day 150). Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant due to the endpoint evaluations occurring at Day 120 and Day 210.

PROTOCOL SUMMARY, Main Criteria for Inclusion and Exclusion. Inclusion Criteria, criteria 9, c and 10

Section 4.4. Inclusion Criteria, criteria 9, c

#### Replace:

- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion

Protocol clarification.


# Section Description of Changes

and 10

10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after

With:

treatment completion

- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus
     52 weeks
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus **52 weeks**

PROTOCOL SUMMARY, Main Criteria for Inclusion and Exclusion, Exclusion Criteria criterion 2 Replace:

2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE)

With:

Section 4.5, Exclusion Criteria, criterion 2

2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic **sclerosis**, or vasculitis not related to SLE)

# PROTOCOL SUMMARY,

Statistical Considerations, Paragraph 2 Add:

Two analyses are planned: 1) an interim analysis to select the POC dose based on the MAD data, and 2) a final analysis at study completion. Additionally, DMC safety analyses will be performed for each MAD cohort and throughout the POC to monitor patient safety as described in the DMC charter. An additional analysis may be performed for the MAD portion of the study when all MAD patients have completed the safety follow-up, or withdrawn from the study, and prior to the final analysis. Data from the POC part of the study will be excluded from this additional analysis.

Replace:

Section 1.2.2.3, Clinical Studies, Paragraph 2

PK data from the SAD study demonstrates BOS161721 has an extended t<sub>1/2</sub> (provisional single dose data indicates this to be approximately 42-46 days) which supports evaluation of monthly dosing.

With:

Final PK data from the SAD study demonstrates BOS161721 has a mean  $t_{1/2}$  ranging from 80 to 87 days for doses of  $\geq$  30 mg in healthy subjects.

Protocol

clarification.

Rationale

Protocol clarification; text added to clarify that additional analysis would allow for flexibility if sponsor wanted to add an IA to review MAD only data.

Updated to reflect that terminal elimination half-life (t½) is due to a full Healthy Volunteer Single Ascending Dose dataset.


| Description of Changes | Rationale |
|---|---|
| Replace: This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD portion (see Section 3.1.1.1). | Respective added section to be referenced. |
| With: | |
| This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD portion (see Section 3.1.2.1 for the chosen POC dose and justification). | |
| Delete: Based on the limited Phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed. | Updated to<br>reflect that all of<br>the data is now<br>acquired and<br>'limited' no<br>longer applies;<br>there were no<br>changes to the<br>safety results. |
| Delete: Based on the limited Phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed. | Updated to reflect that all of the data is now acquired and 'limited' no longer applies; there were no changes to the safety results. |
| Delete: Based on the limited Phase 1 SAD study (BOS161721-01), infections in subjects who received BOS161721 was not observed. | Updated to<br>reflect that all of<br>the data is now<br>acquired and<br>'limited' no<br>longer applies;<br>there were no<br>changes to the<br>safety results. |
| | Replace: This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD portion (see Section 3.1.1.1). With: This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD portion (see Section 3.1.2.1 for the chosen POC dose and justification). Delete: Based on the limited Phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed. Delete: Based on the limited Phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed. |


#### Protocol Date and Version: 23 January 2019; V5.0 Section **Description of Changes** Rationale Updated to Section 1.2.5.5, Delete: reflect that all of Malignancy Based on the limited Phase 1 SAD study (BOS161721-01), malignancy the data is now acquired and in subjects who received BOS161721 was not observed. 'limited' no longer applies; there were no changes to the safety results. Section 1.2.5.6, Delete: Updated to Hepatic Function reflect that all of Abnormality, the data is now Based on the limited Phase 1 SAD study (BOS161721-01), hepatic Paragraph 2 function abnormality in subjects who received BOS161721 was not acquired and 'limited' no observed. longer applies; there were no changes to the safety results. Section 1.2.5.7, Replace: Protocol Failure of clarification; Vaccination, The effect of BOS161721 was evaluated in *in vivo* single dose studies text added for Paragraph 2 in Cynomolgus monkey in which the animals received vaccination to specificity. T-cell dependent KLH antigen to stimulate a TDAR. These in vivo studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen; however, it is worth noting that BOS161721 administration did not produce any remarkable changes in anti-KLH antibody data for IgM, IgG1, IgG3, and IgG4 or anti-tetanus toxoid (TT) antibody data for IgM, IgG, IgG1, or IgE during the dosing phase in the same study. With: The effect of BOS161721 was evaluated in *in vivo* single dose studies in Cynomolgus monkey in which the animals received vaccination to T-cell dependent KLH antigen to stimulate a TDAR. These in vivo studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen in a dose-dependent fashion; however, BOS161721 administration did not affect anti-tetanus toxoid antibody data for IgM, IgG, IgG1, or immunoglobulin E (IgE) during the dosing phase in the same study. Replace:

Section 3.1.2.1, BOS161721 POC Dose Selection and Justification

3.1.2.1 BOS161721 Dose

The optimal dose is chosen based on MAD Phase 1b safety, tolerability, immunogenicity, and PK and PD data. The dose will be Added text for POC dose and justification.


#### Section Description of Changes

Rationale

communicated by a letter to site investigators participating in the POC Phase 2 portion, and to the IRB/IEC.

With:

#### 3.1.2.1 BOS161721 POC Dose Selection and Justification

The dose for the POC portion of the study is 120 mg administered SC monthly (a total of 7 doses). The rationale for the BOS161721-02 Phase 2 POC dose selection was based on cumulative safety, tolerability, immunogenicity, PK, and PD data available from an interim analysis (IA) performed during the MAD Phase 1b portion of the trial.

The data cut-off for this IA occurred on CC and and included all 6 patients and 7 doses from Cohort 1 (20 mg), 12 patients and 6 doses from Cohort 2 (60 mg), and 12 patients and 4 doses from Cohort 3 (120 mg).

The safety analysis focused on incidence and severity of all AEs, SAEs, and pre-determined adverse events of special interest (see Section 6.2.2.6). The DMC and designated unblinded Boston Pharmaceuticals team met on CCI and did not identify any untoward safety signals at any BOS161721 dose levels.

Because there were no safety, tolerability, or immunogenicity trends observed at the time of the IA, the Phase 2 POC dose selection was made based on available PK and PD data. pSTAT3 levels were assessed as the primary PD biomarker of IL-21R signaling levels. This is because IL-21R signaling, upon IL-21 binding, initially involves phosphorylation of JAK1/JAK3 which dissociate from the receptor complex, and phosphorylate STAT3 which translocates to the nucleus and drives IL-21-regulated gene expression.



The 120 mg dose will be communicated to site investigators participating in the POC Phase 2 portion, and to Institutional Review Boards (IRBs) and the Independent Ethics Committee (IEC).

Section 3.1.2.2, POC Study Design, Paragraph 2 Delete:

As in the MAD part of the study, each patient in the POC portion may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Section 3.4). Dose selection will be based on the DMC and sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD portion of 30

Remove text to reduce redundancy with Section 3.1.2.1


#### Section Description of Changes

#### Rationale

#### patients treated with BOS161721/placebo.

#### Section 3.2,

Randomization and blinding, Paragraph 4

Replace:

An independent biostatistician not otherwise involved on the study will be unblinded and prepare materials for the interim analysis (IA) and the DMC safety reviews.

Added in order to allow for ongoing analysis of the data in the IAs.

With:

An independent biostatistician not otherwise involved on the study will be unblinded and prepare materials for the IA, ad hoc analyses as needed, and the DMC safety reviews.

# Section 3.3, Study Schematic

#### Replace:

Protocol clarification.



#### With:



Section 3.4, Schedule of Assessments, Table 1, Footnote

Add:

| а | Screen*a | Enrollo | | | | Tre | atment- | Period: | Follow- | Up∙o | | | | Safet | Follow | -Upa |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dayso | -28-<br>to-10 | <b>0</b> a | 7¶<br>(±º1)a | 15¶<br>(±3)□ | 30¶<br>(±%)□ | 44¶<br>(±%)¤ | 60¶<br>(±3)¤ | 90¶<br>(±%)¤ | 120¶<br>(±%)□ | 150¶<br>(±%)0 | 180¶<br>(±%)¤ | 187¶<br>(±%)¤ | 195¶<br>(±%)0 | 210¶<br>(±3)¤ | 240¶<br>(±°3)□ | 270¶<br>(±%)¤ |
| Visit-Numbero | 10 | 20 | 0 | 30 | 40 | 5a | 60 | 70 | 80 | <b>9</b> a | 100 | 0 | | 110 | 12a | 130 |
| SLEDAI-2Kho | Χ¤ | Χ¤ | | | Χ¤ | | Xo | Χo | Χ¤ | Χ¤ | Xo | a | D | Χ¤ | Χ¤ | Xα |

h SLEDAI-2K should be done before randomization and

Footnote added for protocol clarification. All subsequent footnotes after 'h' were relettered accordingly.


## Section Description of Changes

Rationale

#### dosing on Day 0 as SLEDAI-2K < 6 is exclusionary.

Section 3.4, Schedule of Assessments, Table 2, Footnote

Add:

■Table 2. → Schedule of Assessments - Phase 2 Proof of Concept (POC)

| 1 | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| •¤ | Screen2° | Enroll□ | | | Tr | eatment | ·Period·I | ollow-u | p⊲ | | | Safe | ty Follo | w-Upa |
| | -28∙ | | 15¶ | 30¶ | 60¶ | 90¶ | 120¶ | 150¶ | 180¶ | 187 <sup>6</sup> | 195 <sup>bq</sup> | 210¶ | 240¶ | 270¶ |
| ■Days¤ | to~l¤ | 0∞ | (±3)∞ | (±3):: | (±3)¤ | (±3)¤ | (±³3)¤ | (±³3)¤ | (±3)≈ | (±3)≈ | (±3)¤ | (±3)∞ | (±°3)≈ | (±3)≈ |
| •Visit·Number∞ | l¤ | 2≈ | 3≈ | <b>4</b> ≈ | 5≈ | 6∞ | 7∷ | 8¤ | 9α | ¤ | ¤ | 10⊲ | 11¤ | 12≈ |

Footnote added for protocol clarification.

Section 3.4, Schedule of Assessments, Table 2, Footnote

Replace:

OPK samples will only be collected at the investigational sites that will be participating in the PK portion of the study.

Footnote added for protocol clarification. All subsequent footnotes after 'b' were relettered accordingly.

With:

PK samples will only be collected at the investigational sites that participate in the PK portion of the study. On PK only days (ie, Day 187 and Day 195 when no laboratory assessments are scheduled) samples will be collected at the investigational sites of the selected countries that participate in the PK portion of the study. Patients not participating in PK are not required to return for investigation site visits on Days 187 and 195.

Section 3.4, Schedule of Assessments, Table 2, Footnote

Add:

Footnote added for protocol clarification.

| •a | Screenso | Enrollo | | | Ti | catment | Period I | ollow-u | p-a | | | Safet | ty Follo | w-Upa |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| • Dayso | -28-<br>to~10 | <b>0</b> a | 15¶<br>(±%)¤ | 30¶<br>(±3)¤ | 60¶<br>(±3)¤ | 90¶<br>(±%)¤ | 120¶<br>(±%)¤ | 150¶<br>(±3)¤ | 180¶<br>(±%)¤ | 187 <sup>65</sup><br>(±%)¤ | 195 <sup>M</sup><br>(±3)0 | 210¶<br>(±%)¤ | 240¶<br>(±%)¤ | 270¶<br>(±3)a |
| ■Visit·Number□ | 10 | 20 | 3α | 40 | 5a | <b>6</b> a | 7a | 8a | 90 | 0 | -0 | 10a | 110 | 12a |
| EFFICACY-ASSESSME | NTSo . | 0 99 1 | 0 10 | | | | | | | | | | | |
| SLEDAI-2K¤ | Xo | Xio | 0 | Χ¤ | Χ¤ | Χo | Χ¤ | X¤ | Χ¤ | D | | Χ¤ | Χ¤ | Χ¤ |

SLEDAI-2K should be done before randomization and dosing on Day 0 as SLEDAI-2K < 6 is exclusionary.

Section 3.4, Schedule of Assessments, Table 2, Predose and Postdose PK Window rows Delete:

| 0 | Screen | Enrolla | | | T | reatmen | Period | Follow-t | pro: | | | Safet | y Follov | w Upo |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| - Dayso | -28-<br>to~10 | 00 | 15¶<br>(±%)o | 30¶<br>(±%)o | 60¶<br>(±%)o | 90¶<br>(±%)¤ | 120¶<br>(±%)a | 150¶<br>(±°3)¤ | 180¶<br>(±3)o | 187#¶<br>(±°3)o | 195°¶<br>(±°3)¤ | 210¶<br>(±%)o | 240¶<br>(±%)o | 2704<br>(±°3) |
| · Visit Numbero | 10 | 20 | 3n | 40 | 5a | <b>6</b> a | 7a | Sa. | 90 | 0 | 0 | 100 | 110 | 12a |
| PK·Labs* | | | | | | | | | | | | | | |
| Predose□ | 0 | Xo | п | Xo | Xo | Χ¤ | Xo | Xo | Xo | п | а | D | | п |
| Predose PK-Window□ | п | 60m□ | | ±-340 | 6-2d0 | #-340 | #-3d0 | ±340 | #-340 | | 10 | | | п |
| Postdose□ | | | X¤ | | - 13 | | | | Ξ. | X□ | X□ | X | Χ¤ | Xo |
| Predose PK-Window□ | π | | ±-340 | п | D. | | - 5 | - 12 | n | ±-3d□ | 4-3d0 | ±-3d0 | 6-340 | ±-24 |

Removed Predose and Postdose PK Window rows to reduce redundancy as these are the same as visit window rows. Repetitive text removed.

Section 4.4, Inclusion Criteria, criterion 7, b, item ii Delete:

Replace:

ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in ≥ 1 joint, (observed or throughout history), with some loss of functional range of movements which lead to some loss of functional range of motion as manifested by effects on instrumental ADLs such as:

Section 4.6.1,

Revised to reduce


#### **Section**

#### **Description of Changes**

#### Corticosteroid

#### 4.6.1 Oral Corticosteroid Dose

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day).

After Day 0 (after initiation of study therapy), no up-titration above 10 mg/day is allowed except for up to 1 CS burst for increased disease activity.

Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits.

- Once a patient has received the first dose of study drug, prednisone (or prednisone equivalent) may be tapered down at the discretion of the investigator.
  - o Tapering is allowed after randomization except within 60 days of the primary (Day 210) and secondary (Day 120) endpoint assessments. Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant.

A maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed during the study between Day 0 and Day 60, according to the following:

- An oral CS "burst" between Day 0 and Day 60; (an increase of ≤ 40 mg/day of prednisone or equivalent), which must be tapered down to a maximum of 10 mg/day within 2 weeks of initiation of the "burst"
  - Alternatively, a single intramuscular (IM) dose of methylprednisolone (40 mg or equivalent) is permitted
  - o The course of the oral CS "burst" is not permitted to extend beyond Day 60

Treatment with inhalational CS therapy (eg, for asthma), or by any other route, is allowed. Other concomitant medications for SLE need to be taken at stable doses as per the inclusion criteria (Section 4.4).

#### With:

#### 4.6.1 Corticosteroid

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment

Rationale

redundancy and improve clarity. Text revised to clarify the meaning of "any other route" and added to address the use of CS for non-SLE conditions. Text regarding other medications not applicable to CS were removed.


## Section Description of Changes

and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day).

Tapering of steroids during the course of the study will be highly encouraged and should be evaluated at the protocol permitted visits (Day 0 through Day 60 and Day 120 through Day 150). Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant due to the endpoint evaluations occurring at Day 120 and Day 210.

- Once a patient has received the first dose of study drug (after Day 0), prednisone (or prednisone equivalent) dose is highly encouraged to continue tapering down as appropriate. The investigator should evaluate the prednisone dose at each visit and make the decision, within the protocol allowed windows.
  - Exception: Between Day 60 and Day 120, and between Day 150 and Day 210 (ie, within 60 days of primary and secondary endpoint assessments), oral CS doses must be held constant.

**After Day 0 (first dose of study drug), a** maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed between Day 0 and Day 60, according to the following:

- The oral CS dose is allowed to increase to ≤ 40 mg/day of prednisone or equivalent, which must be tapered down to ≤ 10 mg/day within 2 weeks of initiation of the "burst"
  - Alternatively, a single intramuscular (IM) dose of methylprednisolone (40 mg or equivalent) is permitted
  - No increase of oral CS above baseline is permitted beyond Day 60

Treatment with inhalational CS therapy (eg, for asthma), or by any other route, but systemic administration, is allowed.

Treatment with intra-articular or intravenous CS is prohibited during the course of the study.

Section 4.7.2, Contraception, Paragraphs 1, 2, and 5 Replace:

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion.

Protocol clarification.

Rationale


#### Section Description of Changes

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion.

Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing.

With:

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks, due to the mean terminal ½ life of the study drug.

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks, due to the mean terminal ½ life of the study drug.

Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, **WOCBP** must still undergo pregnancy testing.

#### Section 5.1, Screening

Add:

Protocol clarification.

Rationale

- Laboratory evaluations (non-fasting):
  - o FSH (postmenopausal women under age 55 years)

Section 6.2.2.5, Seriousness of Adverse Events Delete:

Revised for clarity.

Text added 1) to

clarify that basal

cell carcinoma

associated with

suppression, but

is not a

neoplasia

immune

• Is another important medical event (see below)

Section 6.2.2.6, Adverse Events of Special Interest Replace:

- 4. Malignancy
- Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, and disseminated tuberculosis

With:

- 4. Malignancy (not including basal cell carcinoma or squamous cell carcinoma of skin)
- Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, disseminated herpes simplex, disseminated tuberculosis, Aspergillus sp., Candida albicans, Coccidioides immitis, Cryptococcus neoformans, Cytomegalovirus, Histoplasma capsulatum, Isospora belli, and Polyomavirus JC polyomavirus

rather secondary to sun exposure and 2) to clarify specific opportunistic infections of special interest in this study.

Section 6.2.2.6.4, Malignancy, Add:

Revised to align with text for


| Section | Description of Changes | Rationale |
|---|---|---|
| Paragraph 2 | After the first dose of study drug, when there is a decision to biopsy a potentially malignant tumor, lymph node, or other tissue (with the exception of suspected basal cell/squamous cell), the investigator and/or consultant(s) should contact the sponsor clinicians or designee to discuss the issue and any decisions as soon as possible. Basal cell carcinoma or squamous cell carcinoma of skin is not considered an AE of special interest. | AEs of special interest. |
| Section 6.2.2.6.5,<br>Special Infections | Replace: Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, shingles, disseminated herpes simplex, or disseminated tuberculosis will be recorded as AEs of special interest. | Revised to align<br>with text for<br>AEs of special<br>interest. |
| | With: | |
| | Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, disseminated herpes simplex, disseminated tuberculosis, Aspergillus sp., Candida albicans, Coccidioides immitis, Cryptococcus neoformans, Cytomegalovirus, Histoplasma capsulatum, Isospora belli, or Polyomavirus JC polyomavirus will be recorded as AEs of special interest. | |
| Section 8, Statistics | <ul> <li>An additional analysis may be performed for the MAD portion of the study when all MAD patients have completed the safety follow-up or withdrawn from the study, and prior to final analysis. Data from the POC part of the study will be excluded from this additional analysis.</li> </ul> | Analysis added<br>to allow the<br>sponsor to<br>perform another<br>interim<br>evaluation of the<br>MAD only data<br>after all subjects<br>complete or |
| Section 8.2.3, Primary Efficacy Endpoint(s) | Delete: Patients that received prohibited medications or unallowable CS usage as described in Section 4.6 will be considered "medication failures" and will be treated as non-responders for the primary efficacy analysis. Patients that received an allowable CS burst but having missing data at Day 210 will considered a medication failure and will be treated as non-responders for the primary efficacy analysis. The determination of medication failures will be reviewed using blinded data and finalized prior to unblinding. | discontinue if wanted. Correction of error in previous version; text is not applicable to the primary efficacy analysis. |
| Appendix 1, Names of<br>Study Personnel,<br>Central Laboratory | Add: PPD | Protocol clarification. |
| | PPD | |


# Section Description of Changes

# Industriepark Zwijnaarde 3b B-9052 Gent, Belgium Replace:

## Appendix 3

| Medication | Dose Equivalence |
|--------------------|------------------|
| Prednisone | 20 mg |
| Cortisone | 100 mg |
| Hydrocortisone | 80 mg |
| Prednisolone | 20 mg |
| Methylprednisolone | 16 mg |
| Triamcinolone | 16 mg |
| Budesonide | 4 mg |
| Dexamethasone | 3 mg |
| Bethamethasone | 2.4 mg |

#### Rationale

Revised to clarify 1:1 equivalence to prednisone.

#### With:

| Medication | Prednisone Dose Equivalence |
|--------------------|-----------------------------|
| Prednisone | 1 mg |
| Cortisone | 5 mg |
| Hydrocortisone | 4 mg |
| Prednisolone | 1 mg |
| Methylprednisolone | <b>0.8</b> mg |
| Triamcinolone | <b>0.8</b> mg |
| Budesonide | <b>0.25</b> mg |
| Dexamethasone | <b>0.16</b> mg |
| Bethamethasone | <b>0.16</b> mg |

#### Appendix 5, Paragraph 1

Replace:



With:



# Appendix 5, bullet b, item ii

Delete:



Protocol clarification.

Protocol clarification.




# A RANDOMIZED DOUBLE-BLIND PHASE 1b/2 COMBINED STAGGERED MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF LIMITED STANDARD OF CARE

**SPONSOR** Boston Pharmaceuticals, Inc.

55 Cambridge Parkway, Suite 400

Cambridge, MA 02142

United States of America (USA)

INVESTIGATIONAL COMPOUND: BOS161721

PROTOCOL NUMBER: BOS161721-02

PHASE Phase 1b/2

INVESTIGATIONAL NEW DRUG (IND) 131796

**NUMBER:** 


**VERSION NUMBER:** V4.0 (Amendment 3)

**VERSION DATE:** 27 July 2018


## CLINICAL PROTOCOL APPROVAL FORM

| Protocol Title: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care | |
|---|---|
| Study Number: BOS161721-02 | |
| Version | Date |
| Original Protocol | 06 October 2017 |
| Protocol Version 2.0 (Amendment 1) | 14 November 2017 |
| Protocol Version 3.0 (Amendment 2) | 21 March 2018 |
| Protocol Version 4.0 (Amendment 3) | 27 July 2018 |

This study protocol was subject to critical review and has been approved by sponsor. The information contained in this protocol is consistent with:

- The current risk-benefit evaluation of the investigational product.
- The moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (APPENDIX 2), and principles of Good Clinical Practices (GCP) as described in 21 Code of Federal Regulations (CFR) parts 50, 54, 56 and 312 and according to applicable local requirements.

The investigator will be supplied with details of any significant or new findings, including adverse events, relating to treatment with the investigational product.

I agree with these statements and indicate my approval by signature for this protocol:

| Name and Title | Signature and Date |
|---------------------------------------------------------|--------------------|
| DDD MD NID | |
| PPD , MD, PhD<br>Chief Medical Officer | |
| Boston Pharmaceuticals | |
| PPD , MD, FACR | |
| Vice President, Clinical Development | |
| Boston Pharmaceuticals | |
| DDD | |
| PPD Clinical Operations Lead | |
| Boston Pharmaceuticals | |
| PPD , MD, PhD | |
| Vice President, Clinical Development and Safety Officer | |
| Boston Pharmaceuticals | |


#### BOS161721-02

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

#### CONFIDENTIALITY AND INVESTIGATOR STATEMENT

The information contained in this protocol and all other information relevant to BOS161721 are the confidential and proprietary information of Boston Pharmaceuticals, Inc., and except as may be required by federal, state, or local laws or regulation, may not be disclosed to others without prior written permission of Boston Pharmaceuticals, Inc.

I have read the protocol (Version 4.0, dated 27 July 2018), including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described. I will conduct this study as outlined herein, in accordance with the regulations stated in the Federal Code of Regulations for Good Clinical Practices and International Council for Harmonisation (ICH) guidelines, and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and any amendments, and access to all information provided by Boston Pharmaceuticals, Inc., or specified designees. I will discuss the material with them to ensure that they are fully informed about BOS161721 and the study.

| Principal Investigator Name (printed) | | Signature |
|---------------------------------------|-------------|-----------|
| Date | Site Number | |


# PROTOCOL SUMMARY

| Title: | A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care |
|---|---|
| Indication | Adults with moderately to severely active SLE |
| Background and Rationale | SLE is a chronic systemic autoimmune disease with considerable heterogeneity in clinical manifestations and disease course. There is evidence that B- and T-cells are critical to the development of the disease, and that T-cell-derived cytokines such as interleukin-21 (IL-21) are involved in the SLE-associated inflammatory pathological response. |
| | BOS161721 is a humanized immunoglobulin G1 (IgG1) triple mutation monoclonal antibody (mAb) intended to have an extended terminal elimination half-life (t <sub>1/2</sub> ) that selectively binds to and neutralizes IL-21, which acts on multiple cell types that drive inflammation and autoimmunity. In vivo, BOS161721 inhibits T-cell dependent antigen responses of B-cells and is being developed as a potential treatment for adults with moderately to severely active SLE. |
| | Nonclinical studies have evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), pharmacokinetics (PK), and immunogenicity of BOS161721 administered intravenously (IV) and subcutaneously (SC). The no observed adverse effect level (NOAEL) in Cynomolgus monkeys was determined to be 100 mg/kg (SC and IV), the highest dose tested. There were no injection site reactions in animals dosed subcutaneously. |
| | In a Phase 1 single ascending dose (SAD) study, BOS161721 was administered IV and SC to healthy male and female adult subjects. This double-blind, placebo-controlled study evaluated 8 ascending dose levels (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) for safety, tolerability, PK, PD and immunogenicity. Overall, there were no clinically significant safety or tolerability findings from this study. |
| | Results from the Phase 1 SAD study informed the dose regimens used for the multiple ascending doses (MAD) Phase 1b portion of this trial. The MAD portion will involve 3 cohorts. The Phase 2 portion will be a proof of concept (POC) part, where dose selection will be based on the data monitoring committee (DMC) and sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD portion of 30 patients treated with BOS161721/placebo. The purpose of the study is to establish a safe and effective dosage for adult patients with moderately to severely active SLE. |


# Objectives and Endpoints:

# MAD Phase 1b

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | ENDI ORVIS |
| • | Cafatri Endmainta |
| To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose. | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness</li> <li>Injection site reactions</li> <li>Columbia Suicide Severity Rating Scale (C-SSRS)</li> <li>12-lead electrocardiograms (ECGs) parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> <li>Clinical laboratory results and change from baseline</li> <li>Physical examinations changes from baseline</li> <li>Anti-drug antibodies (ADAs)</li> <li>Study drug exposure/compliance</li> </ul> |
| Secondary | study utug enposite compilation |
| To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PD effects in patients with mild to moderate SLE. | <ul> <li>Pharmacokinetic Endpoints</li> <li>BOS161721 concentration by visit and time point</li> <li>Maximum observed concentration (C<sub>max</sub>), first time to maximum concentration (T<sub>max</sub>), area under the concentration-time curve (AUC), t½, systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>)</li> <li>Pharmacodynamic Endpoints</li> <li>Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype</li> <li>Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit</li> <li>Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit</li> </ul> |

## Exploratory





# **POC Phase 2**

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To demonstrate a superior effect of<br>BOS161721 at the chosen dose<br>compared with placebo for<br>response on the SLE Responder<br>Index 4 (SRI-4) | Primary Efficacy Endpoint The proportion of patients with a SRI-4 response at Day 210 (see Section 6.3.4.1) |
| Secondary | |
| To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment | <ul> <li>The proportion of patients with: <ul> <li>SRI-4 response at each visit</li> <li>SRI-5 and SRI-6 response at each visit (Section 6.3.4.2)</li> <li>a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210</li> <li>new BILAG A flare or &gt; 1 BILAG B flares relative to baseline through Day 210</li> <li>PGA worsening</li> <li>a BICLA response</li> <li>a CLASI response</li> <li>medication failures</li> </ul> </li> <li>Results and changes from baseline in: <ul> <li>CLASI</li> <li>swollen and tender joints ACR-28</li> <li>SLEDAI-2K</li> <li>SLICC/ACR damage index</li> </ul> </li> <li>Time to medication failure</li> <li>Duration of longest SRI-4 response</li> <li>Time to first SRI-4 response</li> <li>Time to BILAG A flare or &gt; 1 BILAG B flare compared to baseline through Day 210</li> </ul> |
| Safety | |
| To assess safety and tolerability of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness</li> <li>Injection site reactions</li> <li>C-SSRS</li> <li>12-lead ECGs parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> <li>Clinical laboratory results and change from</li> </ul> |




#### **Study Design:**

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of multiple SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, eligible patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly. The trial will consist of 2 double-blinded portions: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

The MAD Phase 1b portion of the study design will consist of 3 cohorts, with Cohort 1 containing 6 patients, where 5 of these patients will receive BOS161721 (active), and 1 will receive placebo. Cohorts 2 and 3 will each contain 12 patients, including 9 active and 3 placebo patients. Dose selection for each cohort is based on 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. Each of the 3 doses (20, 60, and 120 mg) selected for the MAD portion are projected not to exceed the mean exposure of that achieved in the SAD study following the single 240 mg SC dose. Each patient may receive a total of


7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

The MAD portion design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after the DMC evaluates the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after the DMC evaluation of the safety and tolerability data from Cohort 2 and Cohort 1. Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. This dose will not exceed doses tested during the MAD portion.

For the POC portion, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio. As in the MAD portion, each patient in the POC portion may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 60. Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits. Tapering may occur after randomization except within 60 days of the primary (Day 210) and secondary (Day 120) endpoint assessments. Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant.

DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.


# Main Criteria for Inclusion and Exclusion

#### **Inclusion Criteria:**

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion OR Lupus nephritis as the sole clinical criterion in the presence of antinuclear antibodies [ANA] or anti- double-stranded deoxyribonucleic acid [dsDNA] antibodies), either sequentially or simultaneously
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
  - c. C3 or C4 levels below normal as determined by the central lab
- 5. At screening, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA,


decreased complement, thrombocytopenia, and leukopenia

- ii. Points from lupus headache and organic brain syndrome will also be excluded
- 7. Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 4.4

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization)
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion
- 10. Men who are sexually active with WOCBP must agree to follow


instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion

11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

#### **Exclusion Criteria**

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary


- a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count < 350/μL at screening
- 16. Platelets < 50,000/mm<sup>3</sup> (50  $\times$  10<sup>9</sup>/L) or < 35,000/ mm<sup>3</sup> (35  $\times$  10<sup>9</sup>/L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation
- 20. Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) > 2 × the upper limit of normal (ULN) at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK) > 3.0  $\times$  ULN at screening unless related to lupus myositis
- 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic mAb (eg, IgG protein) or molecules made of components of


#### mAbs

- 25. History substance and/or alcohol abuse, or dependence within the past 1 year, at the investigator's judgment
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 on the C-SSRS
- 31. Current or pending incarceration
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness

# Statistical Considerations

Below is a summary of the statistical methods. Further details can be found in Section 8.

Two analyses are planned: 1) an interim analysis to select the POC dose based on the MAD data, and 2) a final analysis at study completion. Additionally, DMC safety analyses will be performed for each MAD cohort and throughout the POC to monitor patient safety as described in the DMC charter.

Unless stated otherwise, statistical testing will only be performed on the POC data and will be done using 2-sided overall alpha of 0.10. Data will be summarized descriptively by treatment and overall for each study phase. For the MAD portion, BOS161721 will be summarized overall and by each dose level and placebo patients from each cohort will be combined.

The descriptive summaries for the categorical data will include number and percentage. The descriptive summaries for the continuous data will include number, mean, median, standard deviations (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, median, and maximum. Counts, medians, 25<sup>th</sup> and 75<sup>th</sup> percentiles,


and standard error will be presented for time-to-event data.

All safety analyses will be performed using the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. All efficacy analyses will be performed using the full analysis set (FAS), defined as all patients who receive at least 1 dose of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. Select efficacy analyses may also be performed on the per protocol (PP) set.

Binary efficacy endpoints, including the primary efficacy endpoint, will be assessed via Pearson's chi-squared analysis.

Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) when applicable, adjusting for the baseline value. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test.

Adverse event data will be coded to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be summarized, based on coded terms, using frequency and percentage of patients. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters, will be summarized at each individual visit.


# **TABLE OF CONTENTS**

| CLINICAL PROTOCOL APPROVAL FORM | 2 |
|----------------------------------------------------|----|
| CONFIDENTIALITY AND INVESTIGATOR STATEMENT | 3 |
| PROTOCOL SUMMARY | 4 |
| TABLE OF CONTENTS | 16 |
| LIST OF IN-TEXT TABLES | 19 |
| LIST OF IN-TEXT FIGURES | 19 |
| LIST OF ABBREVIATIONS | 20 |
| 1. INTRODUCTION AND RATIONALE | 24 |
| 1.1 Indication | 24 |
| 1.2 Background and Rationale | 24 |
| 1.2.1 Overview of the Disease State | 24 |
| 1.2.2 BOS161721 Development | 24 |
| 1.2.2.1 Interleukin-21 | 25 |
| 1.2.2.2 Preclinical Studies | 26 |
| 1.2.2.3 Clinical Studies | 27 |
| 1.2.3 Study Dose Selection | 28 |
| 1.2.4 Risk-Benefit Assessment | 29 |
| 1.2.5 Potential Risks | 30 |
| 1.2.5.1 Anaphylaxis and Serious Allergic Reactions | 31 |
| 1.2.5.2 Injection Site Reactions | 31 |
| 1.2.5.3 Immune Complex Disease | 31 |
| 1.2.5.4 Infections | 32 |
| 1.2.5.5 Malignancy | 32 |
| 1.2.5.6 Hepatic Function Abnormality | 33 |
| 1.2.5.7 Failure of Vaccination | 33 |
| 1.2.5.8 Potential for Drug-Drug Interactions | 34 |
| 1.2.5.9 Potential Risk to Fetal Development | 34 |
| 2 STUDY OBJECTIVES AND ENDPOINTS | 34 |
| 2.1 Phase 1b Multiple Ascending Dose | 34 |
| 2.2 Phase 2 Proof of Concept | 36 |
| 3 STUDY PLAN | 37 |
| 3.1 Study Design | 37 |
| 3.1.1 Multiple Ascending Dose Phase 1b | 37 |
| Dose Escalation for the MAD Portion | 38 |
| Dose Limiting Toxicity (DLT) | 38 |
| 3.1.1.3 DMC Recommendations | 39 |
| 3.1.2 POC Phase 2 | 39 |
| 3.1.2.1 BOS161721 Dose | 39 |

| Clinical Study Protocol: BOS161721-02 | |
|-----------------------------------------------|---|
| Protocol Date and Version: 27 July 2018; V4.0 | ) |

| 3.1.2.2 | POC Study Design | 39 |
|---|---|---|
| 3.2 | Randomization and Blinding | |
| 3.3 | Study Schematic | 41 |
| 3.4 | Schedule of Assessments | 42 |
| 3.5 | End of Study | 51 |
| 4 P | OPULATION | 51 |
| 4.1 | Participant Recruitment | 51 |
| 4.2 | Number of Patients | 51 |
| 4.3 | Patient Screening | 51 |
| 4.4 | Inclusion Criteria | 51 |
| 4.5 | Exclusion Criteria | 54 |
| 4.6 | Concomitant Medications | 56 |
| 4.6.1 | Oral Corticosteroid Dose | 56 |
| 4.6.2 | Other Prohibited and/or Restricted Treatments | 57 |
| 4.7 | Women of Childbearing Potential | 57 |
| 4.7.1 | Determination of Menopause | 58 |
| 4.7.2 | Contraception | 58 |
| 4.8 | Deviation from Inclusion/Exclusion Criteria | 59 |
| 4.8.1 | Patient Withdrawal and Replacement | 59 |
| 5 S | TUDY PROCEDURES | 59 |
| 5.1 | Screening | 59 |
| 5.1.1 | Retesting During Screening Period. | 60 |
| 5.2 | <u> </u> | |
| 5.3 | 5.3 Treatment Period/Follow-Up Visits | |
| 5.4 | 5.4 Safety Follow-Up Visits | |
| 5.5 | 5.5 Premature Discontinuation | |
| 6 A | ASSESSMENTS | 64 |
| 6.1 | Medical History, Demographic and Other Baseline Information | |
| 6.2 | Safety Assessments | 64 |
| 6.2.1 | Laboratory Assessments | 64 |
| 6.2.1. | Pregnancy testing | 66 |
| 6.2.1.2 | 2 Tuberculosis Screening | 66 |
| 6.2.2 | Adverse Events | 67 |
| 6.2.2. | 1 Definitions | 67 |
| 6.2.2.2 | 2 Recording of Adverse Events | 67 |
| 6.2.2. | 3 Severity of Adverse Events | 67 |
| 6.2.2.4 Causality of Adverse Events 6 | | |
| 6.2.2.: | | |
| 6.2.2. | 1 | |
| 6.2.2. | 7 Reporting of Adverse Events | 72 |
| 6.2.2. | 8 Follow Up of Adverse Events | 74 |

| Clinical Study Protocol: BOS161721-02 | |
|-----------------------------------------------|---|
| Protocol Date and Version: 27 July 2018; V4.0 | 0 |

| 6.2.3 | Vital Signs | 74 |
|---------|--------------------------------------------------------------|----|
| 6.2.4 | 12-Lead Electrocardiograms | 74 |
| 6.2.5 | Physical Examinations | 74 |
| 6.2.6 | C-SSRS | 75 |
| 6.2.7 | Injection Site Reactions | 75 |
| 6.2.8 | Immunogenicity | 75 |
| 6.3 | Efficacy Assessments | 76 |
| 6.3.1 | SLEDAI-2K | 76 |
| 6.3.2 | BILAG 2004 | 76 |
| 6.3.3 | PGA of Disease Activity | 76 |
| 6.3.4 | Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response | 77 |
| 6.3.4.1 | | |
| 6.3.4.2 | SRI-5 and SRI-6 Response | 77 |
| 6.3.4.3 | BICLA Response | 77 |
| 6.3.5 | CLASI Response | 77 |
| 6.3.6 | ACR-28 Joint Count | 77 |
| 6.4 | Other Variables | 78 |
| 6.4.1 | SLICC/ACR Damage Index | 78 |
| 6.4.2 | PROs | 78 |
| 6.5 | Pharmacokinetic Assessments | 78 |
| 6.6 | Pharmacodynamic Assessments | 78 |
| 6.7 | Pharmacokinetic/Pharmacodynamic Relationship | 79 |
| 6.8 | Protocol Deviations | 79 |
| 7 S | TUDY DRUG MANAGEMENT | 79 |
| 7.1 | Description | 79 |
| 7.1.1 | Formulation | 79 |
| 7.1.2 | Storage | 79 |
| 7.2 | Packaging and Shipment | 79 |
| 7.3 | Dose and Administration | 79 |
| 7.4 | Accountability | 80 |
| 7.5 | Prohibited Concomitant Therapy | 80 |
| 7.6 | Compliance | 80 |
| 8 S | TATISTICS | 80 |
| 8.1 | Sample Size | 81 |
| 8.2 | Statistical Methods | 82 |
| 8.2.1 | Analysis Populations | 82 |
| 8.2.2 | Demographics and Baseline Characteristics | 82 |
| 8.2.3 | Primary Efficacy Endpoint(s) | 82 |
| 8.2.4 | Secondary Efficacy Endpoint(s) | 83 |
| 8.2.5 | Analysis of Safety | 83 |
| 8.2.5.1 | Safety Analysis | 83 |

| Clinical Study Protocol: BO | OS161721-02 |
|-----------------------------|--------------------|

| 8.2.6 | Pharmacokinetic and Pharmacodynamic Data | 83 |
|---|---|---|
| 8.2.6.1 Analysis of Pharmacokinetic Data | | |
| 3.2.6.2 Analysis of Pharmacodynamic Data | | |
| 8.2.6.3 | Population Pharmacokinetic Analysis or PK/PD Modeling | 84 |
| 8.3 Inter | rim Analysis and Power | 84 |
| 9 ETHIC | ETHICS AND RESPONSIBILITIES | |
| 9.1 Goo | .1 Good Clinical Practice | |
| 9.2 DM | | |
| 9.3 Insti | tutional Review Board/Independent Ethics Committee | 85 |
| 9.4 Info | rmed Consent | 85 |
| 9.5 Reco | ords Management | 86 |
| 9.6 Sour | rce Documentation | 86 |
| 9.7 Stud | ly Files and Record Retention. | 87 |
| | TNG AND MONITORING | |
| | DMENTS | |
| | Y REPORT AND PUBLICATIONS | |
| 13 STUDY DISCONTINUATION | | |
| | DENTIALITY | |
| | ENCES | |
| | NDICES | |
| APPENDIX 1 NAMES OF STUDY PERSONNEL | | |
| APPENDIX | | |
| APPENDIX | | |
| APPENDIX | | |
| APPENDIX | , | |
| APPENDIX | | |
| APPENDIX | 7 PROTOCOL SUMMARY OF CHANGES | 102 |
| | LIST OF IN-TEXT TABLES | |
| Table 1. | Schedule of Assessments - Phase 1b - Multiple Ascending Dose | 42 |
| Table 2. | Schedule of Assessments - Phase 2 Proof of Concept (POC) | |
| Table 3. | Laboratory Tests | |
| Table 4. | Causality Definitions | |
| | LIST OF IN-TEXT FIGURES | |
| Figure 1. | Individual pSTAT3 C <sub>min</sub> Levels Versus Dose | 29 |
| Figure 2. | • | |
| -8 | igure 2. Study Diagram for Mild Flage 10 and 1 OC I have 2 | |


BOS161721

Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 27 July 2018; V4.0

# LIST OF ABBREVIATIONS

ACR American College of Rheumatology

ADA anti-drug antibody
AE adverse event

AIDS acquired immune deficiency syndrome

ALT alanine aminotransferase
ANA antinuclear antibodies
ANC absolute neutrophil count
ANOVA analysis of variance

ANCOVA analysis of covariance
APL antiphospholipid

AST aspartate aminotransferase

AUC area under the concentration-time curve

AZA azathioprine

BICLA BILAG-based Composite Lupus Assessment

BILAG British Isles Lupus Assessment Group

BP blood pressure BUN blood urea nitrogen

BW body weight
C complement
CS corticosteroids

C-SSRS Columbia Suicide Severity Rating Scale

CD cluster of differentiation

CK creatine kinase

C<sub>L</sub> systematic clearance

CLASI Cutaneous Lupus Erythematosus Area and Severity Index

C<sub>max</sub> maximum plasma concentration

CMH Cochran-Mantel-Haenszel

CS corticosteroids

CSR clinical study report
DILI drug-induced liver injury
DLT dose-limiting toxicity

DMC data monitoring committee

dsDNA double-stranded deoxyribonucleic acid

ECG electrocardiogram EOT end of treatment

eCRF electronic case report form

F female

CCI

FAS full analysis set


Fc fragment crystallizable

FDA Food and Drug Administration FSH follicle stimulating hormone

GCP Good Clinical Practice

eGFR estimated glomerular filtration rate

GLP Good Laboratory Practice

GWAS genome-wide association studies

γc gamma chain HBV hepatitis B virus

hCG human chorionic gonadotropin

HCl hydrochloride HCV hepatitis C virus

HIV human immunodeficiency virus

HR heart rate

HRT hormone replacement therapy

IA interim analysis

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonization

IEC Independent Ethics Committee

Ig immunoglobulin IL interleukin

IL-21R interleukin 21 receptor

IM intramuscular INFy interferon gamma

INR International Normalized Ratio IRB Institutional Review Board

IUD intrauterine device

IV intravenous

IVRS interactive voice response system

JAK Janus kinase kg kilogram

KLH keyhole limpet hemocyanin LOCF last observation carried forward

M male

mAb monoclonal antibody
MAD multiple ascending dose

MAPK mitogen-activated protein kinase

MedDRA Medical Dictionary of Regulatory Activities

MS multiple sclerosis MTX methotrexate


BOS161721 Boston Pharmaceuticals, Inc.


NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NIAID/FAAN National Institute of Allergy and Infectious Diseases/Food Allergy and

Anaphylaxis Network

NK natural killer

NOAEL no observed adverse event level

NO nitric oxide
OTC over-the-counter
PD pharmacodynamics
PEF peak expiratory flow

PGA Physician's Global Assessment

PK pharmacokinetics
POC proof of concept
PP per protocol

PR (interval) from onset of the p-wave to the end of the r-wave

pSS primary Sjögren's syndrome

pSTAT3 phosphorylated signal transducer and activator of transcription 3

PT preferred term

QRS (interval) from the onset of the q-wave to the end of the s-wave
QT (interval) from onset of the QRS complex to the end of the T wave
QTcF QT interval corrected for heart rate using Fridericia's formula

QFT-G QuantiFERON-TB Gold In-Tube

RA rheumatoid arthritis

RR (interval) from the onset of the r-wave to the onset of the next consecutive r-

wave

SAD single ascending dose SAE serious adverse event SAP statistical analysis plan

SC subcutaneous

SDMT safety data monitoring board

CCI

SLE systemic lupus erythematosus
SLEDAI-2K SLE Disease Activity Index 2000

SLICC Systemic Lupus International Collaborating Clinics

Sm Smith

SOC system organ class
SRI-4 SLE Responder Index 4
SRI-5 SLE Responder Index 5
SRI-6 SLE Responder Index 6
SS safety analysis set

SSA Sjögren syndrome-A (Ro) SSB Sjögren syndrome-B (La)


BOS161721 Boston Pharmaceuticals, Inc.


STAT3 signal transducer and activator of transcription 3 SUSAR suspected unexpected serious adverse reaction

terminal elimination half-life

TB tuberculosis

TDAR T-cell dependent antibody response

Tfh T-follicular helper

Th T-helper
TK toxicokinetics

T<sub>max</sub> first time to maximum concentration

Treg regulatory T-cell TT tetanus toxoid

ULN upper limit of normal

US United States

Vd volume of distribution

WBC white blood cell

WHO World Health Organization
WOCBP women of childbearing potential

YTE triple mutation


# 1. INTRODUCTION AND RATIONALE

#### 1.1 Indication

BOS161721 is a humanized monoclonal antibody (mAb), which binds to and inhibits interleukin-21 (IL-21) bioactivity, and is being developed for the treatment of moderately to severely active systemic lupus erythematosus (SLE) in adults.

# 1.2 Background and Rationale

#### 1.2.1 Overview of the Disease State

SLE is a chronic inflammatory autoimmune disease that has variable manifestations in multiple organ systems and follows a relapsing and remitting course. The disease process includes abnormal immune responses mediated by tissue-binding autoantibodies and immune complex deposition, giving rise to tissue damage often resulting in end organ disease and even mortality. Survival of SLE has improved due to earlier detection, improved overall medical care, and standardized SLE treatment with corticosteroids (CS), immunosuppressants, and cytotoxic agents. However, some of the morbidity in patients with SLE is related to its treatment. Comparison of early and late outcomes in patients with SLE demonstrate that death in early disease is most commonly due to infections and active SLE causing multi-system organ damage, while thromboses were the most common cause of death during later disease.<sup>2</sup>

The reported prevalence of SLE in the United States (US) is 20 to 70 cases per 100,000 people.<sup>3</sup> More than 90% of cases of SLE occur in women, frequently starting at childbearing age. Women of color are disproportionately affected by SLE. This suggests multiple genetic and environmental factors are at play. Accordingly, a multifactorial view of the immunopathogenesis of SLE suggests more than 1 area of interest, including breach in central tolerance in the adaptive arm of the immune system, peripheral amplification of the autoimmune response by the innate immune system, and local processes in the target organ that facilitate end-organ disease.<sup>4</sup>

# **1.2.2 BOS161721 Development**

Boston Pharmaceuticals is developing BOS161721 for the treatment of SLE. BOS161721 is a humanized immunoglobulin G1 (IgG1) mAb with extended half-life directed against human IL-21.

Murine mAb 19E3, the progenitor of BOS161721, was generated using mouse hybridoma technology. 19E3 has subpicomolar (pM) affinity to human IL-21 and was selected for its potent neutralization of IL-21 bioactivity. BOS161721 was generated by the humanization of mAb 19E3 where its complementarity-determining regions were grafted onto a human IgG1 kappa backbone. The fragment crystallizable (Fc) portion of BOS161721 contains a YTE (M252Y/S254T/T256E triple mutation) in the constant domain of the IgG1 heavy chain that was introduced into the parental molecule, 19E3, intended to prolong the in vivo terminal elimination half-life (t<sub>1/2</sub>) of the mAb.<sup>5</sup> Thus, BOS161721 retains sub-pM binding to IL-21 and prevents IL-21 from binding to the IL-21 receptor (IL-21R), inhibiting IL-21 bioactivity.


BOS161721 binds to human IL-21 and Cynomolgus monkey IL-21, which are highly homologous, and neutralizes the bioactivity of both. BOS161721 is specific for IL-21 as it does not bind to or inhibit the other gamma-chain (γc) family of cytokines, and acts to specifically neutralize the IL-21 pathway. In *in vitro* studies, BOS161721 inhibited downstream IL-21-induced signaling, IL-21-induced plasma cell differentiation, and IL-21-induced natural killer (NK) cell activation. In *in vivo* studies, BOS161721 significantly inhibited the T-cell dependent antibody response (TDAR) to immunization with a protein antigen as well as B-cell expansion following a second protein antigen immunization in Cynomolgus monkeys.

#### 1.2.2.1 Interleukin-21

IL-21 is an inflammatory cytokine, which belongs to a family of cytokines that also includes IL-2, IL-4, IL-7, IL-9, and IL-15, all of which bind to private receptors in complex with the common cytokine receptor yc. 6 Most cytokines in this family are critically important for both the maintenance and function of T-cell and B-cell responses. IL-21 signals through a receptor complex consisting of its own private receptor, the IL-21R and yc.<sup>6,7</sup> Engagement of the IL-21R/γc complex leads to the activation of several signaling pathways, including the Janus kinase/signal transducer and activator of transcription, mitogen-activated protein kinase (MAPK) and phosphoinositide 3-kinase pathways. 8 IL-21 is produced mainly by T-cells and NK T-cells, but neutrophils have also been reported to produce IL-21.9,10 The IL-21R is expressed on a broad array of cell types, including B-cells, T-cells, NK-cells, macrophages and dendritic cells, as well as other hematopoietic and nonhematopoietic cells such as fibroblasts, keratinocytes, and intestinal epithelial cells. 9,11 Activation of signal transducer and activator of transcription 3 (STAT3) via phosphorylation is critical in regulating human B-cell responses to IL-21<sup>12</sup>; phosphorylated STAT3 (pSTAT3) forms a homodimer, which translocates to the nucleus where it initiates transcription of the IL-21 gene, forming an autocrine loop for IL-21 production via STAT3 phosphorylation. <sup>13</sup> In addition, IL-21 has been shown to upregulate expression of its own receptor 14 and induces an autocrine feedback loop. 15

IL-21 modulates various aspects of immune function. It promotes cluster of differentiation 4 (CD4+) T-cell differentiation and promotes the generation of T-helper (Th)17<sup>16</sup> and T-follicular helper (Tfh) cells. <sup>15,17</sup> In mice, IL-21 has been shown to regulate the balance between Th17 and regulatory T-cell (Treg), in that it increases Th17, while inhibiting Treg differentiation. <sup>18</sup> Less is understood with regards to human Tregs, although IL-21 has been reported to counteract Treg suppression of human effector T-cells <sup>19</sup> and blockade of IL-21 promotes Treg generation in a murine model of graft versus host disease induced by human T-cells. <sup>20</sup> IL-21 upregulates CD8+ T-cell and NK-cell expansion and cytolytic activity by increasing granzyme B and perforin. <sup>21,22</sup> IL-21 also has been reported to increase granzyme B in plasmacytoid dendritic cells and B-cells resulting in inhibition of T-cell responses. <sup>23,24</sup> IL-21 also has a variety of effects on nonhematopoietic cells, such as stromal cells and induces inflammation through matrix metalloproteinase release by gut intestinal fibroblasts. <sup>25</sup>

One principal non-redundant role of IL-21 is the promotion of B-cell activation, differentiation, or death during humoral immune responses. <sup>14</sup> Furthermore, increased IL-21 production is characteristic of several autoimmune diseases and is likely to contribute to autoantibody production as well as pathologic features of autoimmune disease. <sup>26</sup> The critical role of IL-21 in promoting humoral and other immune responses makes it an important focus of potential


therapeutic interventions in conditions characterized by overproduction of pathogenic autoantibodies. IL-21 production by Tfh cells in humans is believed to play a major role in driving the autoantibody production through its role in plasma cell differentiation. Importantly, Tfh cell populations are expanded in patients with autoimmune diseases such as lupus, bullous pemphigoid, rheumatoid arthritis (RA) and primary Sjögren's syndrome (pSS) and have been reported to correlate with IL-21 levels, autoantibodies, and disease severity. <sup>26,27,28,29</sup> Furthermore, loss of number and functionality of Tregs has been associated with autoimmune diseases such as SLE and giant cell arteritis, which IL-21 is expected to modulate. <sup>30,31</sup> Thus, neutralization of IL-21 in settings of autoimmunity is expected to impact several cell populations believed to be involved in the pathogenesis of autoimmune disorders including SLE.

BOS161721 selectively binds IL-21 with high affinity to neutralize IL-21, and due to its pleiotropic nature, neutralization of IL-21 is expected to impact several cell populations believed to be involved in the pathogenesis of SLE. Importantly, patients with SLE have elevated IL-21 plasma levels that correlate with the severity of the disease. Recently, genome-wide association studies (GWAS) have provided convincing evidence that the chromosomal 4q 27 region harbors the IL-21 genes and is associated with chronic inflammatory disorders, including SLE.<sup>29</sup>

#### 1.2.2.2 Preclinical Studies

The pharmacokinetics (PK) of BOS161721 were characterized following single-dose intravenous (IV) administration of BOS161721 (0.01 to 30 mg/kg) in male Cynomolgus monkeys or repeat, every 2 weeks IV administration (15 to 100 mg/kg) and subcutaneous (SC) administration (50 mg/kg) in male and female Cynomolgus monkeys. Systemic exposure was approximately dose-proportional within the tested dose range. SC bioavailability was determined to be 64.3%.

Two single-dose (IV) non-good laboratory practice (GLP) studies conducted in Cynomolgus monkeys evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), and immunogenicity of BOS161721. Following a single IV administration (slow bolus), there were no BOS161721-related adverse changes, resulting in a no-observed-adverse-effect-level (NOAEL) value of 30 mg/kg, the highest dose tested among 2 studies.

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) administration for 3 months (a total of 7 doses).




An additional GLP, repeat-dose toxicity study was conducted in Cynomolgus monkeys (4 males and 4 females per dose group) following every 2 weeks (Q2W) administration by SC (10, 30, and 100 mg/kg) injection for a total of 14 doses.



#### 1.2.2.3 Clinical Studies

BOS161721-01 was a double-blind, Phase 1, single ascending dose (SAD) study to assess the safety, PK, and PD of BOS161721 in healthy subjects. The primary objective of the study was to characterize the safety and tolerability of IV and SC SADs of BOS161721 in an otherwise healthy subject population without concomitant illnesses, immune abnormalities, or concomitant medications. Secondary objectives included characterization of the PK and immunogenicity of BOS161721, and exploratory objectives included the evaluation of the effect of BOS161721 on TDAR to keyhole limpet hemocyanin (KLH) (primary and secondary immunizations) in healthy subjects, the effects of BOS161721 on plasma levels of IL-21 (free and bound), and the evaluation of the effect of BOS161721 on IL-21 gene expression (via gene signature) in blood. This study consisted of 8 cohorts. Subjects were randomized in a 3:1 ratio (BOS161721: placebo) and received either a single dose of BOS161721 (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) or placebo, with safety follow-up. For the first cohort, after the first 2 subjects were dosed (1 active and 1 placebo), there was a minimum gap of 48 hours before the remaining subjects from that cohort were dosed, to allow for an initial review of any emerging safety and tolerability data. For all cohorts, escalation to the next dose was not


sooner than 8 days after all the subjects in the prior cohort had been dosed and were based on a review of at least 7 days of safety and tolerability data by the Safety Data Monitoring Team (SDMT).

Blood samples were collected at every in-house study visit for BOS161721 concentration determinations. Blood samples were also collected for determination of IL-21 plasma levels (free and total). Safety was assessed based on the occurrence of treatment-emergent AEs, hepatic function abnormality, and acute and delayed hypersensitivity reactions. Other safety variables included ECGs, vital signs (blood pressure [BP], heart rate, and temperature), safety laboratory assessments, blood sampling for ADAs, total IgG and immunoglobulin M (IgM) levels, CD4+ count, and full and targeted physical examinations. Overall, there were no clinically significant findings from this study. Adverse events reported as related to the study drug, particularly infections, were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. There was 1 serious adverse event (SAE; death due to pulmonary embolism) that occurred 127 days after a single administration of 240 mg SC dose of BOS161721. The causality of this single SAE was not attributed to study drug and further information can be found in the Investigator's Brochure. PK data from the SAD study demonstrates BOS161721 has an extended t<sub>1/2</sub> (provisional single dose data indicates this to be approximately 42-46 days) which supports evaluation of monthly dosing.

#### 1.2.3 Study Dose Selection

Doses have been selected for the multiple ascending dose (MAD) Phase 1b portion based on a 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01); the SDMT reviewed the blinded safety data from subjects for each dose cohort (8 cohorts, evaluating 1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg), along with the accumulated safety and available PK/PD data from all subjects in the previous dose cohorts, to make a decision on whether to proceed to the next higher dose level, repeat a dose level, or stop dose escalation. Overall, there were no clinically significant safety or tolerability findings from this study.

Based on the Day-90 interim cut of the PK and biomarker data in the BOS161721-01 study, the recommended doses for evaluation in the MAD portion of this study are 20, 60, and 120 mg SC monthly. This dose recommendation is supported by evidence of linear PK with BOS161721 resulting in a median first time to maximum concentration (T<sub>max</sub>) of 6 days and an apparent terminal half-life of 44 days. Furthermore, pSTAT3 suppression, a marker of IL-21 target engagement, follows a similar time course of the mAb levels, with maximal and sustained suppression apparent with doses greater than 30 mg SC (Figure 1).


pSTAT3 cmin (percent pSTAT3+ lymphocytes, stimulated) 60 pSTAT3 cmin Route IV SC 20 100 0 50 150 200 250 Dose (mg)

Figure 1. Individual pSTAT3 C<sub>min</sub> Levels Versus Dose

IV = intravenous, pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SC = subcutaneous

All doses selected for the MAD portion are projected not to exceed the mean exposure of that achieved following the highest single dose of 240 mg SC administered in the Phase 1 SAD study. Cohort 1 will include randomized treatment to the 20 mg dose. Based on the staggered study design, the data monitoring committee (DMC) will perform a scheduled review of safety data and sequentially consider dose escalation for Cohorts 2 and 3. In addition, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the proof of concept (POC) Phase 2 portion. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD portion (see Section 3.1.1.1).

#### 1.2.4 Risk-Benefit Assessment

The available preclinical data on BOS161721, the findings in clinical study BOS161721-01, and existing clinical information on IL-21 inhibitors suggest that the present clinical study has an acceptable risk-benefit ratio. In this study, the risk-benefit assessment of BOS161721 in adult patients with moderately to severely active SLE will be ongoing, with step-wise evaluations during the staggered MAD portion. The DMC used in this study is charged with assessing such actions in light of an acceptable benefit-risk profile for BOS161721 as an anti-IL-21 mAb.


Formal DMC monitoring meetings will occur as described in the DMC Charter. Two weeks after Cohort 1 has received a second dose of study drug, the DMC will evaluate the safety and tolerability data from Cohort 1 to determine the recommended dose for Cohort 2. Two weeks after 8 patients in Cohort 2 receive a second dose, the DMC will determine if dose escalation to Cohort 3 can proceed. Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 during the MAD part of study. Thereafter, DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter. With the agreement of the DMC and sponsor, this schedule may be modified depending on the rate of patient accrual. Additional details can be found in the DMC Charter.

The benefit of participation for all patients in this study is close monitoring of their medical condition and safety of their treatment. Those randomized to the active treatment arm may potentially experience improvement in their SLE disease. Those randomized to the placebo (in combination with standard of care) arm are not expected to obtain any additional benefit, beyond those of their background treatment, though close monitoring of their medical condition and safety may itself be associated with improving their SLE.

#### 1.2.5 Potential Risks

Potential risks based on the mechanism of action of BOS161721 include infections, risks associated with the administration of any foreign protein or biologic agent, including injection site reaction, anaphylaxis, serious allergic reaction, and development of ADAs. ADAs could result in immune complex disease (with manifestations such as arthralgias, serum-sickness, and vasculitis), or altered BOS161721 levels or activity. Further details can be found in the current Investigator's Brochure (IB) for BOS161721, which contains comprehensive toxicology, preclinical and clinical information on BOS161721.

Two investigational drug products are considered to be in the same pharmacological class as BOS161721 based on interruption of signaling through the IL-21 signaling pathway. No potential risk generalizable across the class has been observed with these investigational products. Based on the clinical Phase 1 SAD study (BOS161721-01), AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs.

The majority of IgG elimination occurs via intracellular catabolism, following fluid-phase or receptor-mediated endocytosis. This type of endocytosis and elimination is a form of target-mediated disposition where the interaction of the drug and its pharmacological target (eg, a target receptor) serves as a significant contributor to the kinetics of antibody distribution and elimination. Renal elimination, which is a primary pathway of clearance of small-molecule drugs, is relatively unimportant for IgG, as its large size prevents efficient filtration through the glomerulus. Secretion into the bile is an important pathway of elimination of IgA antibodies, but this route is not a significant contributor to the elimination of IgG antibodies. Thus, risk to renal and hepatic systems due to metabolism of BOS161721 is low.<sup>33</sup>


# 1.2.5.1 Anaphylaxis and Serious Allergic Reactions

As with the administration of any foreign protein and/or other biological agents, acute hypersensitivity reactions, including acute anaphylactic/hypersensitivity, severe allergic, and anaphylactoid reactions may follow infusion of mAbs and can be caused by various mechanisms. These acute hypersensitivity reactions may be severe and result in death.

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria,<sup>34</sup> and are discussed in Section 6.2.2.6.1.

Based on the limited Phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed.

Patients with a known history of allergy or severe hypersensitivity reaction to any component of BOS161721 formulation or patients with a history of anaphylaxis to any other biological therapy such as mAbs will be excluded from studies with BOS161721. In addition, appropriate drugs and medical equipment to treat acute hypotensive, bronchoconstrictive, or anaphylactic reactions will be immediately available at the unit and study personnel will be trained to recognize and treat these reactions.

#### 1.2.5.2 Injection Site Reactions

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC for 3 months (a total of 7 doses). There were no injection site reactions in animals dosed subcutaneously. Further, there were no reports of injection site reactions in the 26-week GLP toxicology study in Cynomolgus monkeys.

Based on the Phase 1 SAD study (BOS161721-01), incidence of injection site reactions in subjects who received BOS161721 was similar to placebo.

Patients will be monitored for local injection site reactions in this study. See Section 6.2.7.

#### 1.2.5.3 Immune Complex Disease

The potential risk of immune complex disease for BOS161721 is theoretical, based on the known risks associated with mAbs. The administration of a mAb can result in the formation of ADAs. Administration of the mAb in the presence of ADA may result in the formation of circulating antibody-antigen complexes potentially resulting in altered BOS161721 levels or activity or deposition of the complexes in microvasculature. Complement is frequently involved in the latter setting, and the breakdown products of complement attract polymorphonuclear leukocytes to the site of deposition where they can provoke local tissue damage through specific or nonspecific release of enzymes. Two of the more common end-organ targets are the blood vessels (vasculitis) and kidney (nephritis). These clinical manifestations represent immune complex disease or Type III hypersensitivity. Although BOS161721 is a humanized mAb, ADAs may develop; however, the likelihood of occurrence of immune complex disease with BOS161721 is low. The findings of immune complex disease are typically reversible when mAb administration stops and the antibody-antigen complexes are cleared from the body.


Based on the limited Phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed.

#### 1 2 5 4 Infections

BOS161721 is expected to diminish the activity of T-cell, B-cell and NK-cell lines. Like other medications modulating immune response, BOS161721 may increase the potential risk for infection, including serious infections. IL-21 produced by CD4+ Th cells is required to sustain the anti-viral function of CD8+ T-cells against chronic viral infections. Nonclinical evidence suggests that the risk of chronic viral infection recurrence or increased severity may occur with IL-21 inhibition.<sup>35</sup>

These conditions will be fully characterized with clinical descriptions and routine laboratory and/or specialty testing and treated where indicated with appropriate local standard of care.

Patients with a history of opportunistic infection, including recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years, or any other underlying pathology predisposing to serious infection, are excluded from studies with BOS161721 (for further details please refer to the current IB for BOS161721).

Patients will be assessed for hepatitis B, and C, and HIV-1/2 combination, at screening.

#### <u>Cryptosporidium Infection</u>

Cryptosporidium infection was noted in patients with an IL-21 receptor loss-of-function gene mutation and similar findings of cryptosporidium infection have been observed in immunosuppressed liver transplant and human immunodeficiency virus patients. Since BOS161721 is expected to diminish the immunosurveillance activity of T-cell, B-cell, and NK-cell lines, a similar risk is biologically plausible with prolonged exposure to BOS161721.

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells,<sup>37</sup> patients with a CD4+ count < 500 cell/mm³ were excluded from the Phase 1 SAD study (BOS161721-01), and CD4 + < 350 cells/mm³ will be excluded from the MAD/POC parts of the study. Patients exposed to investigational product who develop diarrhea during the course of the study should immediately undergo an assessment for opportunistic infection including stool for ova and parasites and stool examination for cryptosporidium. Positive cryptosporidium in stool sample at screening is an exclusion. Treatment by the investigator where indicated should be guided by findings and be consistent with local standard of care.

Based on the limited Phase 1 SAD study (BOS161721-01), infections in subjects who received BOS161721 was not observed.

#### 1.2.5.5 Malignancy

The stimulatory effect of IL-21 on NK cells and CD8+ T-cells suggests the cytokine may have anti-tumor activity. Nonclinical studies have demonstrated significant anti-tumor effects of IL-21 in a number of tumor models. IL-21 therapy of human metastatic melanoma and renal cell carcinoma has demonstrated POC with significant increases in levels of perforin, granzyme B,


and interferon gamma (IFN $\gamma$ ) expression in CD8+ T-cells and NK T-cells. Clinical response has been limited in these generally unmanageable diseases.

The impact of treatment with anti-IL-21 therapy on the development or growth of malignancies is not known; however, as with other immunomodulatory biologic agents, treatment with BOS161721 may result in an increase in the risk of malignancies. NK cell suppression by IL-21 neutralization may represent a biological mechanism for a potential risk for malignancy. Patients with a history or current diagnosis of cancer within the past 5 years, with the exception of non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy, are excluded from the study.

Based on the limited Phase 1 SAD study (BOS161721-01), malignancy in subjects who received BOS161721 was not observed.

# 1.2.5.6 Hepatic Function Abnormality

There is no substantial evidence suggesting BOS161721 is associated with liver function abnormality. However, as a precaution, patients with a history of abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST >  $2 \times \text{upper limit of normal [ULN]}$ ; total bilirubin >  $1.5 \times \text{[ULN]}$  and judged by the investigator to be clinically significant) were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from this trial. Patients with a positive hepatitis B or C test or a history of alcohol dependence will also be excluded.

Based on the limited Phase 1 SAD study (BOS161721-01), hepatic function abnormality in subjects who received BOS161721 was not observed.

#### 1.2.5.7 Failure of Vaccination

IL-21 is a key cytokine in development of B-cells into immunoglobulin-secreting plasma cells. Abnormal signaling through the IL-21R/Janus Kinase (JAK)3/signal transducer and activator of transcription (STAT3) pathway leads to defective humoral immune responses to both T-dependent and T-independent antigens and impairs the establishment of long-lasting B-cell memory. Abnormal signaling through the pathway has been related to decreased specific antibody responses following vaccination, and to increased susceptibility to encapsulated bacterial infections.<sup>38</sup>

The effect of BOS161721 was evaluated in in vivo single dose studies in Cynomolgus monkey in which the animals received vaccination to T-cell dependent KLH antigen to stimulate a TDAR. These in vivo studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen; however, it is worth noting that BOS161721 administration did not produce any remarkable changes in anti-KLH antibody data for IgM, IgG1, IgG3, and IgG4 or anti-tetanus toxoid (TT) antibody data for IgM, IgG, IgG1, or IgE during the dosing phase in the same study.


#### 1.2.5.8 Potential for Drug-Drug Interactions

Drug-drug interactions were not evaluated in the Phase 1 SAD study (BOS161721-01), which included only healthy adult subjects. Use of prescription medications (with the exceptions of oral contraceptives), and over-the-counter (OTC) treatments including herbal supplements such as St John's Wort (except multivitamins), in the 2 weeks prior to screening was prohibited in the SAD study.

See Section 4.5 for other specific exclusion criteria which support lowered risk of interactions, and Section 4.6.1 for corticosteroid (CS) dosing. In addition, Section 1.2.5.6 describes considerations for hepatic function for this study.

# 1.2.5.9 Potential Risk to Fetal Development

No data on preclinical reproductive toxicity are available at the time of this study.

# 2 STUDY OBJECTIVES AND ENDPOINTS

This trial has separate objectives and endpoints for the MAD Phase 1b and POC Phase 2 portions of the study. The primary, secondary, and exploratory objectives for each phase, as applicable, are described below with their corresponding endpoints.

# 2.1 Phase 1b Multiple Ascending Dose

| OF | BJECTIVES | ENDPOINTS |
|---|---|---|
| Pr | imary | |
| • | To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose. | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of AEs and SAEs, related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness</li> <li>Injection site reactions</li> <li>Columbia Suicide Severity Rating Scale (C-SSRS)</li> <li>12-lead ECGs parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> <li>Clinical laboratory results and change from baseline</li> <li>Physical examinations changes from baseline</li> <li>ADAs</li> <li>Study drug exposure/compliance</li> </ul> |
| | Secondary | |
| • | To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PD effects in patients with mild to moderate SLE. | Pharmacokinetic Endpoints BOS161721 concentration by visit and time point Maximum observed concentration (C <sub>max</sub> ), T <sub>max</sub> , area under the concentration-time curve (AUC), terminal elimination half-life (t <sub>1/2</sub> ), systematic clearance (C <sub>L</sub> ), volume of distribution (V <sub>d</sub> ) |


# Pharmacodynamic Endpoints Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit **Exploratory** CCI CCI


# 2.2 Phase 2 Proof of Concept

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To demonstrate a superior effect of<br>BOS161721 at the chosen dose compared<br>with placebo for response on the SRI-4 | Primary Efficacy Endpoint The proportion of patients with a SRI-4 response at Day 210 (see Section 6.3.4.1) |
| Secondary | |
| To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment | <ul> <li>The proportion of patients with: <ul> <li>SRI-4 response at each visit</li> <li>SRI-5 and SRI-6 response at each visit (Section 6.3.4.2)</li> <li>a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210</li> <li>new BILAG A flare or &gt; 1 BILAG B flares relative to baseline through Day 210</li> <li>PGA worsening</li> <li>a BICLA response</li> <li>a CLASI response</li> <li>medication failures</li> </ul> </li> <li>Results and changes from baseline in: <ul> <li>CLASI</li> <li>swollen and tender joints ACR-28</li> <li>SLEDAI-2K</li> <li>SLICC/ACR damage index</li> </ul> </li> <li>Time to medication failure</li> <li>Duration of longest SRI-4 response</li> <li>Time to first SRI-4 response</li> <li>Time to BILAG A flare or &gt; 1 BILAG B flare compared to baseline through Day 210</li> </ul> |
| Safety | |
| To assess safety and tolerability of repeat<br>doses of BOS161721 (20, 60, and<br>120 mg) administered SC in adult patients<br>with moderately to severely active SLE<br>on limited background standard of care<br>treatment | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness</li> <li>Injection site reactions</li> <li>C-SSRS</li> <li>12-lead ECGs parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> <li>Clinical laboratory results and change from baseline</li> <li>Physical examinations changes from baseline</li> </ul> |
| | <ul> <li>ADAs</li> <li>Study drug exposure/compliance</li> </ul> |

# **Exploratory**




#### 3 STUDY PLAN

# 3.1 Study Design

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, eligible patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly.

The trial will consist of 2 double-blinded portions: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

SLE disease activity assessment data will be centrally reviewed by medical monitor and sponsor to ensure the scores are clinically meaningful and compliant with specific definition. The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease activity. Further details on the content and methods of data reports by the medical monitor and sponsor will be outlined in the Medical Data Review Plan along with the processes and procedures that will be followed.

# 3.1.1 Multiple Ascending Dose Phase 1b

The MAD portion will consist of 3 cohorts:

• Cohort 1 (20 mg SC) will include 6 patients


- o 5 patients will receive BOS161721 (active group) and 1 patient will receive placebo (placebo group)
- Cohorts 2 (60 mg SC) and 3 (120 mg SC) will include 12 patients each
  - o 9 patients in the active group and 3 in the placebo group

Doses selected for each of the 3 cohorts is based on a 90-day safety, tolerability, PK and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. All doses selected for the MAD part of the study are projected not to exceed the mean exposure of that achieved in the SAD study.

#### 3.1.1.1 Dose Escalation for the MAD Portion

The MAD portion of the study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after the DMC evaluation of the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after the DMC evaluation of the safety and tolerability data from Cohorts 1 and 2. Each cohort will continue at their assigned dose level through their respective 6-month treatment periods (See Study Schematic, Section 3.1). If patients discontinue the study in a cohort prior to adequate safety follow-up, he/she may be replaced.

Criteria for dose escalation are further described in the DMC Charter. See Section 3.1.1.2 for additional details about DLTs.

#### 3.1.1.2 Dose Limiting Toxicity (DLT)

Severity of adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs occurring after study drug administration, which are attributable to the study drug, will be considered DLTs:

#### Hematologic:

- Grade 4 neutropenia
- Grade 3 neutropenic infection
- Grade 3 thrombocytopenia with bleeding
- Grade 4 thrombocytopenia

#### **Non-Hematologic:**

• Grade 3 or above toxicities, persisting after optimal treatment with standard medical therapy (eg. anti-emetics, anti-diarrheals)


• Drug-induced liver injury ([DILI], Hy's Law), as defined in Section 6.2.2.6.3

Investigators should always manage their patients according to their medical judgment which may include interruption of study drug based on the particular clinical circumstances.

# 3.1.1.3 DMC Recommendations

During scheduled meetings, the DMC will review relevant study data for safety or benefit-risk concern. During the MAD part of the study, the DMC may provide the following recommendations to the sponsor:

- Expanding a cohort at a specific dosing level, or repeating a lower dose in a subsequent cohort
- Continuing a dose level for a given cohort
- Escalating a dose level for a subsequent cohort
- Termination of current or previous cohort(s)

Further dosing in a given cohort will be halted if 2 or more DLTs are identified intra- and inter-patients dosed. For the POC portion, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC Phase 2 part of the study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD portion. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available 30 days after the last patient from Cohort 3 receives the third dose. Details are provided in the DMC Charter.

#### **3.1.2 POC Phase 2**

#### 3.1.2.1 BOS161721 Dose

The optimal dose is chosen based on MAD Phase 1b safety, tolerability, immunogenicity, and PK and PD data. The dose will be communicated by a letter to site investigators participating in the POC Phase 2 portion, and to the IRB/IEC.

#### 3.1.2.2 POC Study Design

For the POC part of the study, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio.

As in the MAD part of the study, each patient in the POC portion may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Section 3.4). Dose selection will be based on the DMC and sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD portion of 30 patients treated with BOS161721/placebo.


BOS161721 Boston Pharmaceuticals, Inc.


DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.

# 3.2 Randomization and Blinding

This is a randomized, double-blind study.

Patients meeting all inclusion and exclusion criteria will be centrally randomized to either placebo or BOS161721 using an IWRS according to a randomization list generated by an independent, non-study statistician. Randomization will be performed separately for each study portion and separately for each cohort in the Phase 1b and 2 portions as follows:

| Phase/Cohort | Number of Patients | Randomization Ratio BOS161721:Placebo |
|---|---|---|
| Phase 1b/Cohort 1 | 6 | 5:1 |
| Phase 1b/Cohort 2 | 12 | 3:1 |
| Phase 1b/Cohort 3 | 12 | 3:1 |
| Phase 2 | 156* | 2:1 |

<sup>\*</sup>Additional patients may be enrolled to ensure sufficient numbers of patients are in the full analysis set (FAS).

Eligible patients will be assigned to the study portion which is active at time of enrollment. Similarly, patients in the Phase 1b MAD will be assigned to the cohort which is active. Each patient will be assigned a unique randomization number which will not be reused.

All patients, investigators, and study team participants will be blinded to treatment assignment. An independent biostatistician not otherwise involved on the study will be unblinded and prepare materials for the interim analysis (IA) and the DMC safety reviews. The DMC will review unblinded data during safety reviews and the IA. A limited team at Boston Pharmaceuticals will review unblinded results from the Phase 1b MAD portion during the IA to determine the dose that will be used for the Phase 2 POC portion of the study. Details regarding maintenance of the blinding and content of data reviews will be described in the DMC charter or related study documentation.


BOS161721 Boston Pharmaceuticals, Inc.


# 3.3 Study Schematic

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2



A = active drug (BOS161721); P = placebo


# 3.4 Schedule of Assessments

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | | Tre | eatment | Period | Follow- | Up | | | | Safet | y Follow | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| GENERAL ASSESS | MENTS | | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | | | | | | | | | | | | | | | | |
| criteria | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| SLICC Criteria for<br>SLE | X | | | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>c</sup> | | X | | | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | | X | | X | X | X | X | X | | | | | |
| SAFETY ASSESSM | ENTS | l . | | ı | Į. | | | ı | ı | ı | I. | l. | ı | | | |
| Full physical exam | X | X | | | | | | | | | | | | | | |
| Chest x-ray <sup>d</sup> | X | | | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>e</sup> | X | X | | | X | | | X | | | | | | | | X |
| Injection site reaction assessment | | Xf | X | | X | | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | | X | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>g</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESS | SMENTS | | | | | | | | | | | | | | | |
| BILAG-2004 Index | X | X | | | X | | X | X | X | X | X | | | X | X | X |


 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | | Tro | eatment | Period | Follow- | Up | | | | Safet | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| SLEDAI-2K | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| PGA of disease | 37 | 37 | | | 37 | | 37 | 37 | 37 | 37 | 37 | | | 37 | 37 | 37 |
| activity | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLICC/ACR<br>Damage Index | | X | | | | | | | | | X | | | | | |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| LABORATORY ASS | SESSMEN | TS | | <u> </u> | | • | | | | • | | • | | | • | |
| CD4+ count | X | X | | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments (hematology and | | | | | | | | | | | | | | | | |
| clinical chemistry)h | X | X | | | X | X | X | X | X | X | X | | | X | X | X |
| Coomb's test directi | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | | X | X | X | | X | | | X | | | | | |
| Plasma CCI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Plasma CCI & | | X | | X | X | | X | X | | | X | | | | | |
| Whole blood for leukocyte | | | | | | | | | | | | | | | | |
| immunophenotype | | X | | X | X | | X | X | | | X | | | | | |
| ADA <sup>j</sup> | | X | | X | X | | X | X | | | X | | | | | X |
| $nAb^k$ | | | | | | | | X | | | X | | | | | |
| pSTAT3 <sup>1</sup> | | X | | | X | X | X | X | | | | | | | | |
| CCI | | X | | X | | | | X | | | X | | | | | X |
| CCI | | X | _ | | | | | | | | | | | | | |


Table 1. Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Tre | eatment | Period | Follow- | Up | | | | Safet | y Follow | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | - | 11 | 12 | 13 |
| CCI | X | X | | | X | | X | X | X | X | X | | | $X^{m}$ | X <sup>m</sup> | X <sup>m</sup> |
| CRP | X | | | | | | | X | | | | | | | | X |
| Serum pregnancy<br>test (women) | X | | | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>n</sup> | | X | | | X | | X | X | X | X | X | | | | | X |
| TB test<br>(QuantiFERON-TB<br>Gold In-Tube) <sup>d</sup> | X | | | | | | | | | | | | | | | |
| Serology (hepatitis<br>B and C, HIV-1/2<br>combination) | X | | | | | | | | | | | | | | | |
| Stool sample <sup>o</sup> | X | | | | | | | | | | | | | | | |
| Spot urine for protein/creatinine ratio | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | | X | | X | X | X | X | X | | | X | X | X |


 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Tre | atment | Period | Follow- | Up | | | | Safet | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (±3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| PK Labs | | | | | | | | | | | | | | | | |
| Predose | | X | | | X | | X | X | X | X | X | | | | | |
| Predose PK<br>Window | | 60m | | | ± 3d | | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | | | | | |
| Postdose | | Xp | X | X | X <sup>p</sup> | | | | | | Xp | X | X | X | X | X |
| Postdose PK<br>Window | | 4h ± 30m<br>8h ± 45m<br>24h ± 60m | ± 1d | ± 3d | 4h ± 30m<br>8h ± 45m<br>24h ± 60m | | | | | | 4h ± 30m<br>8h ± 45m<br>24h ± 60m | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CCl ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; d = day; ECG = electrocardiogram; CCl ; FSH = follicle stimulating hormone; h = hour; HR = heart rate; HIV = human immunodeficiency virus;

IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; m = minute; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SAE = serious adverse event; SC = subcutaneous; CC | ; SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; TB = tuberculosis; TDAR = T-cell dependent antigen response.

- <sup>a</sup> Screening assessments will be performed over more than 1 visit.
- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 4.6.1 for further details.
- <sup>c</sup> Randomization should occur after patient eligibility has been confirmed by central eligibility review.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- <sup>e</sup> ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed at 2 hours postdose.
- Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, 187, and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.


 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Tre | atment | Period | Follow- | Up | | | | Safet | y Follow | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) |
| Visit Number | 1 | 2 | - | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | - | | 11 | 12 | 13 |

- Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.
- When clinically indicated for hemolytic anemia.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed (analyzed) if the patient had a positive ADA on Day 90.
- <sup>k</sup> nAb is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90.
- <sup>1</sup> Predose (trough) samples only.
- m Only CCl collected during safety follow-up visits.
- <sup>n</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- Oryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- Postdose samples will be collected at 4, 8, and 24 hours after study drug administration on Days 0, 30, and 180.


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | Tı | reatment | t Period 1 | Follow-u | ıp | | | Safe | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| GENERAL ASSESSMENTS | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| SLICC Criteria for SLE | X | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>c</sup> | | X | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | X | X | X | X | X | X | | | | | |
| SAFETY ASSESSMENTS | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | |
| Chest x-ray <sup>d</sup> | X | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>e</sup> | X | X | | X | | X | | | | | | | | X |
| Injection site reaction | | | | | | | | | | | | | | |
| assessment | | X <sup>f</sup> | | X | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and | | | | | | | | | | | | | | l |
| temperature) <sup>g</sup> | X | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESSMENTS | 1 | | | | | I | 1 | 1 | T | | I | 1 | 1 | |
| BILAG-2004 Index | X | X | | X | X | X | X | X | X | | | X | X | X |
| SLEDAI-2K | X | X | | X | X | X | X | X | X | | | X | X | X |
| PGA | X | X | | X | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | X | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | X | X | X | X | X | X | | | X | X | X |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | T | reatmen | t Period | Follow-u | ıp | | | Safet | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| SLICC/ACR Damage Index | | X | | | | | | | X | | | | | |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |
| LABORATORY ASSESSMENT | S | | | | | | | | | | | | | |
| CD4+ count | X | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments | | | | | | | | | | | | | | |
| (hematology and clinical | | | | | | | | | | | | | | |
| chemistry) <sup>h</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Coomb's test directi | X | X | | X | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | X | X | | X | | | X | | | | | |
| Plasma CC | X | X | | X | X | X | X | X | X | | | X | X | X |
| Plasma CCI & CCI | | X | X | X | | X | | | X | | | | | |
| Whole blood for leukocyte | | *** | 3.7 | *** | | 37 | | | *** | | | | | |
| immunophenotype | | X | X | X | | X | | | X | | | | | |
| ADA <sup>j</sup> | | X | X | X | X | X | | | X | | | | | X |
| nAb <sup>k</sup> | | | | | | X | | | X | | | | | |
| CCI | | X | X | | | X | | | X | | | | | X |
| CCI | | X | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | |
| | X | X | | X | X | X | X | X | X | | | $X^{l}$ | $X^{l}$ | $X^{l}$ |
| CRP | X | | | | | X | | | | | | | | X |
| Serum pregnancy test (women) | X | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>m</sup> | | X | | X | X | X | X | X | X | | | | | X |
| TB test (QuantiFERON-TB Gold In-Tube) <sup>d</sup> | X | | | | | | | | | | | | | |
| Serology (hepatitis B and C,<br>HIV-1/2 combination) | X | | | | | | | | | | | | | |


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | Т | reatmen | t Period | Follow-u | ір | | | Safet | y Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | - | - | 10 | 11 | 12 |
| Stool sample <sup>n</sup> | X | | | | | | | | | | | | | |
| Spot urine for protein/creatinine | | | | | | | | | | | | | | |
| ratio | X | X | | X | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | X | X | X | X | X | X | | | X | X | X |
| PK Labs <sup>o</sup> | | | | | | | | | | | | | | |
| Predose | | X | | X | X | X | X | X | X | | | | | |
| Predose PK Window | | 60m | | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | | | | | |
| Postdose | | | X | | | | | | | X | X | X | X | X |
| Predose PK Window | | | ± 3d | | | | | | | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CC ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; d = day; ECG = electrocardiogram; CC ; FSH = follicle stimulating hormone; h = hour; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; m = minute; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; SAE = serious adverse event; SC = subcutaneous; CC ; SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; TDAR = T-cell dependent antigen response.

- <sup>a</sup> Screening assessments will be performed over more than 1 visit.
- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 4.6.1 for further details.
- Randomization should occur after patient eligibility has been confirmed. The actual randomization procedure can be completed on Day -1 after eligibility confirmation or the morning of Day 0 prior to dosing for logistical purposes.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- e ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed at 2 hours postdose.
- yital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 187 and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC)

| | Screena | Enroll | | | Т | reatmen | t Period | Follow-u | ıp | | | Safet | y Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |

- Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.
- When clinically indicated for hemolytic anemia.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed (analyzed) if the patient had a positive ADA on Day 90.
- <sup>k</sup> nAb is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90.
- Only CCl collected during safety follow-up visits.
- <sup>m</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- <sup>n</sup> Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- <sup>o</sup> PK samples will only be collected at the investigational sites that will be participating in the PK portion of the study.


## 3.5 End of Study

**End of Study (Individual Patient):** A patient is considered at the end of study if he/she has withdrawn, prematurely discontinued, or completed all of the study procedures including the last visit.

**End of Study (End of trial):** The end of the study is defined as the date of the last visit of the last patient in the study globally, or the date of which the last patient withdraws or discontinues if all prior enrolled patients have already completed/withdrawn.

#### 4 POPULATION

# 4.1 Participant Recruitment

Advertisements approved by the IRB, and investigator databases, may be used as recruitment procedures for adult men and women with moderately to severely active SLE.

#### 4.2 Number of Patients

Approximately 186 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD Phase 1b portion, and approximately 156 additional patients will be randomized in the POC Phase 2 portion. Note that approximately 24 dropouts are assumed.

# 4.3 Patient Screening

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Section 3.4]) for this study must be performed between Day -28 and Day -1.

#### 4.4 Inclusion Criteria

Patients who meet the following criteria will be considered eligible to participate in this clinical study:

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1


immunologic criterion or Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously

- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
  - c. C3 or C4 levels below normal as determined by central lab
- 5. At screening, the SLE Disease Activity Index 2000 (SLEDAI-2K) must be ≥ 6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 7. Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - i. "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis in ≥ 2 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living that has been present on several days cumulatively over the past 30 days, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
      - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):


> Ambulation, toileting, grooming- including bathing and dressing; feeding oneself

- ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in ≥ 1 joint, (observed or throughout history), with some loss of functional range of movements which lead to some loss of functional range of motion as manifested by effects on instrumental ADLs such as:
  - Cooking, driving, using the telephone or computer, shopping, cleaning, etc, and has been present on several days over the last 30 days, and is present at the time of the screening visit

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization) (see APPENDIX 3)
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures


#### 4.5 Exclusion Criteria

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed.
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study. (See Section 4.6 for prohibited concomitant medication)
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness


- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count < 350/μL at screening
- 16. Platelets < 50,000/mm³ (50  $\times$  109/L) or < 35,000/ mm³ (35  $\times$  109/L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation<sup>39</sup>:

GFR = ([1 for male] or [0.85 for female]) 
$$\times$$
 (140 – Age)  $\times$  BW / (72  $\times$  Creatinine)

- 20. Serum ALT and/or serum AST > 2  $\times$  ULN at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK)  $> 3.0 \times$  ULN at screening, unless it is related to lupus myositis
- 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (eg, IgG protein) or molecules made of components of monoclonal antibodies
- 25. History substance and/or alcohol abuse or dependence within the past 1 year, at the investigator's judgment
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision)
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer


- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4 or 5 on the C-SSRS
- 31. Current or pending incarceration

32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness

#### 4.6 Concomitant Medications

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Patients should stay on stable regimen of other concomitant medications for the treatment of SLE (eg, analgesics, NSAIDs, statins, ACE inhibitors/ARBs and other antihypertensive drugs), unless changes in these treatments are clinically indicated. Use of any other drugs for non-SLE conditions, including over-the-counter medications and herbal preparations, should remain stable unless change or addition is clinically necessary. Discussion with the medical monitor prior to initiation of new medication is strongly recommended. Any concomitant therapies must be recorded on the eCRF. Prior and concomitant medication use will be recorded for the 30 days prior to screening until the last follow-up visit. In addition, historical treatment for SLE (including immunosuppressant, anti-malarial, corticosteroid, and/or biologic agent) will be recorded for the 48 weeks prior to screening in the eCRF.

#### 4.6.1 Oral Corticosteroid Dose

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day).

After Day 0 (after initiation of study therapy), no up-titration above 10 mg/day is allowed except for up to 1 CS burst for increased disease activity.

Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits.

- Once a patient has received the first dose of study drug, prednisone (or prednisone equivalent) may be tapered down at the discretion of the investigator
  - Tapering is allowed after randomization except within 60 days of the primary (Day 210) and secondary (Day 120) endpoint assessments. Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant.

A maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed during the study between Day 0 and Day 60, according to the following:


• An oral CS "burst" between Day 0 and Day 60; (an increase of ≤ 40 mg/day of prednisone or equivalent), which must be tapered down to a maximum of 10 mg/day within 2 weeks of initiation of the "burst"

- o Alternatively, a single intramuscular (IM) dose of methylprednisolone (40 mg or equivalent) is permitted
- o The course of the oral CS "burst" is not permitted to extend beyond Day 60

Treatment with inhalational CS therapy (eg, for asthma), or by any other route, is allowed. Other concomitant medications for SLE need to be taken at stable doses as per the inclusion criteria (Section 4.4).

#### 4.6.2 Other Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in APPENDIX 4. Medications taken within 30 days prior to screening must be recorded on the eCRF.

- 1. Prior exposure to BOS161721
- 2. Patients who have received treatment with anti-CD20 monoclonal antibodies within 24 weeks of screening; recovery of B cells (CD19+) must be documented (record absolute number of CD19+ B cells)
- 3. Patients who have received treatment with cyclophosphamide within the 24 weeks prior to screening
- 4. Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria within 4 weeks for oral use or 8 weeks for topical use of screening
- 5. Patients who are currently receiving or are scheduled to receive plasmapheresis or lymphapheresis therapy, or have received such therapy within 24 weeks prior to screening
- 6. Patients who have received any live vaccines within 30 days of screening. Note: Furthermore, live vaccines should not be used during the course of the study and within the 2 months following last dose. Other inactivated vaccines such as tetanus, etc, may be used according to local guidelines during treatment period
- 7. Patients who are scheduled or anticipated to have elective surgery during the course of the study
- 8. Initiation of new immunosuppressant or anti-malarial agent is not permitted. Note: Dose reduction or replacement may be allowed due to intolerability or shortage for patients on a stable dose prior to study initiation

# 4.7 Women of Childbearing Potential

WOCBP is defined as any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) and is not postmenopausal.


See Section 4.7.2 for detailed information regarding contraceptive requirements for WOCBP.

### 4.7.1 **Determination of Menopause**

Menopause is defined as at least 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes. Women under the age of 55 years must have a documented serum FSH level > 40 mIU/mL at screening to confirm menopause.

### 4.7.2 Contraception

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion.

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion.

Investigators shall counsel WOCBP and men who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and men who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, patients must agree to the use of 1 method of highly effective contraception from the following:

- Male condoms with spermicide
- Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as 1 of the acceptable methods of contraception since they will not be receiving study drug.
- IUDs, such as ParaGard®
- Vasectomy
- Complete abstinence, defined as complete avoidance of heterosexual intercourse, is an
  acceptable form of contraception. Women who are abstinent while participating in the study
  must continue to have pregnancy tests. Acceptable alternate methods of highly effective
  contraception must be discussed in the event that the patient chooses to forego complete
  abstinence.

Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing.


#### 4.8 Deviation from Inclusion/Exclusion Criteria

Deviation from the inclusion or exclusion criteria will not be allowed. If deviation of inclusion/exclusion criteria is discovered after randomization, the investigator should contact the medical monitor for discussion. A decision will be made whether to allow a patient to continue or withdrawal from the study medication.

See Section 6.8 for additional details.

#### 4.8.1 Patient Withdrawal and Replacement

See Section 5.5 for reasons for removal from the trial. Withdrawn patients may be replaced during the MAD part of the study after discussion between the principal investigator or designee and sponsor.

#### 5 STUDY PROCEDURES

Refer to the eCRF completion guidelines for data collection requirements and documentation of study assessments/procedures.

### 5.1 Screening

Screening will be the same for both the MAD and POC portions of the study.

Screening will take place from Day -28 to Day -1, and assessments may be performed over more than 1 visit. Confirmation that the most current IRB/IEC approved informed consent form (ICF) has been signed must occur before any study-specific screening procedures are performed. Procedures that are part of standard of care are not considered study-specific procedures and may be performed prior to informed consent and used to determine eligibility.

All screened patients will be assigned a unique screening number. The screening number will include a 3-digit site number and a 4-digit sequential number to identify patients from the time of screening. Only eligible patients who are confirmed by central review as meeting the inclusion/exclusion criteria, listed in Section 4.4 and Section 4.5 respectively, will be enrolled in the study. Screened patients who drop out of the clinical study before randomization will be recorded as screen failures. If rescreening occurs, the site will assign a new screening number.

Specific procedures at the screening visit will include:

- Medical history documentation
- Review of inclusion and exclusion criteria
  - o Patient medical records must contain documentation of SLE diagnosis
  - o C-SSRS
- Concomitant medication documentation
- Demographics
- Full physical examination


- Vital signs
- Chest x-ray (a prior x-ray can be used if taken within 12 weeks of screening date)
- Laboratory evaluations (non-fasting):
  - Hematology and clinical chemistry
  - o Serology (Hepatitis B and C; HIV-1/2 combination)
  - o TB test
  - o CRP
  - o Direct Coomb's test (if indicated for hemolytic anemia)
  - o CD4+ count, total IgG and IgM levels, plasma CCl , CCl
  - Serum pregnancy test (WOCBP)
  - o FSH (postmenopausal women)
  - o Spot urine for protein/creatinine ratio
  - Urinalysis
  - Stool sample
- 12-lead ECG
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, Physician's Global Assessment (PGA) of disease activity

Screening procedures are listed in the Schedule of Assessments (Section 3.4), and details are provided in Section 6.

#### **5.1.1** Retesting During Screening Period

A single retesting of laboratory parameters and/or other assessments during the screening period is permitted (in addition to any parameters that require a confirmatory value) only if:

- medically indicated
- there is evidence a laboratory sample was mislabeled, indeterminate, inadequately processed, and/or deteriorated in transit to the central laboratory

Any new result will override the previous result (ie, the most current result prior to randomization) and is the value by which study inclusion/exclusion will be assessed, as it represents the patient's most current clinical state. This will also apply to patients who are being rescreened.

## 5.2 Enrollment/Randomization and Day 0 Treatment

Randomization should occur after patient eligibility for enrollment has been confirmed by the central eligibility review.

Prior to randomization, the study site should confirm that the patient still meets inclusion/exclusion criteria (especially SLE disease activity and treatment). The site will obtain a randomization number when registering the patient in IWRS. All patients will receive


BOS161721 or placebo according to the kit number assigned by the IWRS randomization scheme.

After randomization, procedures include:

- PROs: CCI
- C-SSRS
- Laboratory evaluations (fasting):
  - Hematology and clinical chemistry
  - o Direct Coomb's test (if indicated for hemolytic anemia)
  - o CD4+ count, total IgG and IgM levels, plasma CCl , plasma CCl , whole blood for leukocyte immunophenotype
  - o ADA
  - o pSTAT3 (predose [trough] samples only in Phase 1b)
  - o CCI
  - o CCI
  - o See Table 1 and Table 2 for details of PK sampling in the MAD and POC portions
  - o Urine pregnancy test will be collected on WOCBP prior to study drug administration
  - Spot urine for protein/creatinine ratio
  - o Urinalysis
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Full physical examination
- Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours postdose on Day 0)
- 12-lead ECG (prior to PK blood draw)
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, PGA)
- SLICC/ACR damage index
- Study drug administration:
  - Administration of BOS161721 or placebo will take place on-site, and is discussed in Section 7.3
- Injection site reaction assessment performed at 2 hours postdose

Procedures on Day 0 are listed in the Schedule of Assessments (Section 3.4), and details are provided in Section 6.

All patients who are enrolled, randomized, and receive study drug, or undergo study-specific procedures should reconsent with any updated versions of IRB/IEC approved informed consents during study participation as applicable and per institutional guidelines.


## 5.3 Treatment Period/Follow-Up Visits

The following procedures will be performed as indicated in the Schedule of Assessments (Table 1 and Table 2). See Schedule of Assessment tables for allowable windows for each visit.

- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- PROs: CC
- Urine pregnancy tests will be collected on WOCBP prior to study drug administration
- Injection site reaction assessments will be performed predose
- Direct Coomb's test (if indicated for hemolytic anemia)
- Spot urine for protein to creatinine ratio
- Urinalysis
- · CCI
- Plasma CCI
- PGA, BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, and the CLASI will be completed
- SLICC/ACR Damage Index will be completed at Day 180
- C-SSRS
- ECGs prior to PK blood draw
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies, respectively
- Fasting hematology and chemistry assessments
- The CD4+ count and total IgG and IgM levels
- Plasma CCl & CCl , ADA, and whole blood for leukocyte immunophenotype
- pSTAT3 (predose [trough] samples only Phase 1b)
- nAb will be analyzed by central lab if patient is positive for ADA
- CRP
- · CCI

# 5.4 Safety Follow-Up Visits

Safety follow-up visits will take place at Days 210, 240, and 270. These visits will include the following assessments as indicated in the Schedule of Assessments (Table 1 and Table 2):

- PROs: CC
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Injection site reactions
- Targeted physical examination


- Vital signs (prior to PK blood draw)
- Spot urine for protein/creatinine ratio and urinalysis
- Concomitant medication documentation
- BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, and PGA
- Fasting clinical laboratory assessments (hematology and clinical chemistry)
- Direct Coomb's test (if indicated for hemolytic anemia)
- Plasma CCI
- · CCI
- 12-lead ECG (prior to PK blood draw)
- CRP
- ADA
- CCI
- Urine pregnancy test
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC portions, respectively

#### 5.5 Premature Discontinuation

While patients are encouraged to complete all study evaluations, they may withdraw from the study at any time and for any reason. Every effort will be made to determine why any patient withdraws from the study prematurely. If the patient is unreachable by telephone, a registered letter, at the minimum, should be sent to the patient requesting him/her to contact the clinic.

All patients who withdraw from the study with an ongoing AE or SAE must be followed until the end of study or until the event is resolved or deemed stable, respectively.

If a patient withdraws prematurely after dosing, an end of treatment (EOT) visit should be performed (Day 180) and a last follow-up visit 90 days after dosing should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 5.4).

Patient participation may be terminated prior to completing the study and the reason recorded as follows:

- AE/SAE
- Protocol deviation
- Lost to follow-up
- Patient withdraws consent at their own request
- Investigator decision
- Decision by sponsor (other than AE/SAE, protocol deviation, or lost to follow-up)

Withdrawn patients may be replaced after discussion between the investigator or designee and sponsor.


#### 6 ASSESSMENTS

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances, outside of the control of the investigator, which may make it unfeasible to perform the test. In these cases, the investigator will take all steps necessary to ensure the safety and wellbeing of the patient. When a protocol required test cannot be performed the investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. All protocol violations are entered directly into the eCRFs.

### 6.1 Medical History, Demographic and Other Baseline Information

The medical history comprises:

- General medical history
- Documentation of SLE diagnosis
- Historical medication therapy for SLE

The following demographic information will be recorded:

- Age
- Ethnic origin (Hispanic/Latino or not Hispanic/not Latino)
- Race (White, American Indian/Alaska Native, Asian, Native Hawaiian or other Pacific Islander, Black/African American)
- Height (without shoes, in cm)
- Body weight, without shoes (kg)
- Body mass index (BMI [kg/m²])

Other baseline characteristics will be recorded as follows:

- Concomitant medication documentation (see Section 4.6)
- Status of child bearing potential and contraception

### **6.2** Safety Assessments

#### **6.2.1** Laboratory Assessments

Laboratory tests will be performed at times defined in the Schedule of Assessments (Section 3.4). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

A central laboratory will be used (with the exception of urine pregnancy tests) to ensure accuracy and consistency in test results. Laboratory/analyte results that could unblind the study (ie, biomarker results) will not be reported to investigative sites. Urinalysis will be performed on


BOS161721


midstream, clean catch specimens. Some biomarkers listed above will not be drawn at some sites due to geographical logistical challenges. See the laboratory manual for details.

Endpoint analyses will be based on changes from baseline assessments at Days 120 and 210.

 Table 3.
 Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| Hemoglobin | BUN | рН | Spot urine for protein/creatinine ratio |
| Hematocrit | Creatinine | Glucose (qual) | FSH <sup>b</sup> |
| RBC count | Glucose (fasting) | Protein (qual) | Urine pregnancy test <sup>c</sup> |
| RDW | Calcium | Blood (qual) | QuantiFERON®-TB Gold In-Tube test |
| MCV | Sodium | Ketones | (QFT-G) <sup>d</sup> |
| MCH | Potassium | Nitrites | Serology <sup>d</sup> (Hepatitis B and C; HIV-1/2 |
| MCHC | Chloride | Leukocyte esterase | combination) |
| Platelet count | Total CO <sub>2</sub> (bicarbonate) | Urobilinogen | Stool sample <sup>e</sup> |
| WBC count | AST, ALT | Urine bilirubin | Serum pregnancy test |
| CD4+ count | Total bilirubin | Microscopy <sup>a</sup> | |
| Total neutrophils | Alkaline phosphatase | | |
| (Abs) | Creatine kinase | | |
| Eosinophils (Abs) | Uric acid | | |
| Monocytes (Abs) | Albumin | | |
| Basophils (Abs) | Total cholesterol | | |
| Lymphocytes (Abs) | (fasting) | | |
| | LDL-C (fasting) | | |
| | HDL-C (fasting) | | |
| | Triglycerides (fasting) | | |
| | Total protein | | |
| | PT/INR | | |

| Additional Tests <sup>f</sup><br>(potential Hy's Law) | Immunogenicity, PD and other<br>Biomarker Tests |
|---|---|
| AST, ALT (repeat) | ADA |
| Total bilirubin (repeat) | $nAb^g$ |
| Albumin (repeat) | pSTAT3 (predose [trough] samples |
| Alkaline phosphatase | only in Phase 1b) |
| (repeat) | Total IgG & IgM |
| Direct bilirubin | Plasma CC |
| Indirect bilirubin | Plasma CCI & CCI |
| GGT | Whole blood for leukocyte |
| Prothrombin | immunophenotype |
| time/international | CCI |
| normalized ratio (repeat) | CCI |
| Creatine kinase (repeat) | Antibodies <b>CC</b> |
| ` • · | |
| | CRP |
| | Direct Coomb's testh |

Abbreviations: Abs = absolute; ADA = anti-drug antibody; ALT = alanine aminotransferase;

CCl ; AST = aspartate aminotransferase; BUN = blood urea nitrogen; C = complement; CD4+ = cluster of differentiation 4; CRP = C-reactive protein;

;; FSH = follicle stimulating hormone;


Table 3.Laboratory Tests

adverse event; SC = subcutaneous; CC

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| GGT = gamma-glu | utamyltransferase; HDL-C = | high-density lipoprotein | cholesterol; HIV = human |
| immunodeficiency | virus; IgG = immunoglobuli | in G; IgM = immunoglob | oulin M; INR = international normalized |
| ration; $IL-21 = interpretation$ | erleukin 21; LDL-C = low-de | ensity lipoprotein cholest | erol; MCH = mean corpuscular |
| hemoglobin; MCH | IC = mean corpuscular hemog | globin concentration; MC | CV = Mean corpuscular volume; |
| nAb = neutralizing | g antibody; pSTAT3 = phospl | horylated signal transduc | er and activator of transcription 3; |
| PT = prothrombin | time; qual = qualitative; RBC | C = red blood cell; RDW | = RBC distribution width; SAE = serious |

- a. On all urine samples.
- b. At screening only, in women who are amenorrheic for at least 12 consecutive months and under 55 years old.

: TB = tuberculosis.

- c. For WOCBP.
- d. Screening only.
- e. At screening, and if a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- f. Additional testing for potential Hy's Law cases only (See Section 6.2.2.6.3).
- g. If patient is positive for ADA.
- h. If clinically indicated for hemolytic anemia.

### 6.2.1.1 Pregnancy testing

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, at the last follow up visit day (Day 270) and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures (see Section 5.4) are specified in the Schedule of Assessments (see Section 3.4).

See Section 6.2.2.7.1 for information on reporting of pregnancies as AEs/SAEs during the study.

#### 6.2.1.2 Tuberculosis Screening

During the screening period, it must be determined and documented that a patient does not have evidence of active or latent or inadequately treated TB per the exclusion criteria (Section 4.5). The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).

# 6.2.1.2.1 Mycobacterium Tuberculosis Testing Using QuantiFERON Test<sup>40</sup>

QuantiFERON®-TB Gold In-Tube (QFT-G) is an in vitro diagnostic test using a peptide cocktail simulating ESAT-6, CFP-10, and TB 7.7 proteins to stimulate cells in heparinized whole blood. Detection of INFγ performed by enzyme-linked immunosorbent assay (ELISA) is used to identify in vitro responses to these peptide antigens that are associated with Mycobacterium


tuberculosis infection. QFT-G is an indirect test for M. tuberculosis infection (including disease) and is intended for use in conjunction with risk assessment, radiography and other medical and diagnostic evaluations.

Test results will be reported as positive, negative, or indeterminate. A negative QFT-G test result is required to meet the inclusion criterion. In the case of an indeterminate result, repeat tests should be permitted for the purpose of determining eligibility of patients to enroll in this study. If a repeat test is indeterminate again, the patient is a screen failure. The procedure for using this test and interpreting the results will be described fully in the laboratory manual, which will be provided to investigators.

#### **6.2.2** Adverse Events

#### 6.2.2.1 Definitions

An AE is defined as any untoward medical occurrence experienced by a study patient, whether or not considered drug related by the principal investigator.

AEs are unfavorable changes in a general condition, subjective or objective signs or symptoms, worsening of pre-existing concomitant disease, and clinically significant abnormality in laboratory parameters observed in a patient in the course of a clinical study.

Non-serious SLE manifestations or abnormal laboratory results related to SLE disease activity would not be recorded as AEs unless they meet the definition for SAEs (Section 6.2.2.5).

#### 6.2.2.2 Recording of Adverse Events

AEs should be collected and recorded for each patient from the date of the first dose of study drug until the end of their participation in the study, including the safety follow up period.

AEs may be volunteered spontaneously by the study patient, or discovered by the study staff during physical examinations or by asking an open, nonleading question such as 'How have you been feeling since you were last asked?' All AEs and any required remedial action will be recorded on the Adverse Events eCRF and Safety Adverse Event Form. The details of the AE, date of AE onset, date of AE outcome, and action taken for the AE will be documented together with the principal investigator's assessment of the seriousness of the AE and causal relationship to the study drug and/or the study procedure.

All AEs should be recorded individually, using diagnostic terms where possible. If the diagnosis is not established, individual symptoms may be reported. The AEs will subsequently be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

## 6.2.2.3 Severity of Adverse Events

Each AE will be assessed by the principal investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 criteria. <sup>41</sup> When changes in the severity (grade) of an AE occur more frequently than once a day, the maximum severity for the event should be noted for that day. Any change in severity of signs


and symptoms over a number of days will be captured by recording a new AE, with the amended severity grade and the date (and time, if known) of the change.

### 6.2.2.4 Causality of Adverse Events

The principal investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (Table 4) should be selected based on medical judgment, considering the definitions below and all contributing factors.

**Table 4.** Causality Definitions

| Related | A clinical event, including laboratory test abnormality, occurs in a plausible time relationship to treatment administration and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (dechallenge <sup>a</sup> ) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge <sup>b</sup> procedure if necessary. |
|---|---|
| Unrelated | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative dechallenge and rechallenge information. Typically explained by extraneous factors (eg, concomitant disease, environmental factors, or other drugs or chemicals). |

- <sup>a</sup> Dechallenge: Upon discontinuation of a drug suspected of causing an AE, the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation (positive dechallenge), or the symptoms continue despite withdrawal of the drug (negative dechallenge). Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia).
- Rechallenge: Upon re-administration of a drug suspected of causing an AE in a specific patient in the past, the AE recurs upon exposure (positive rechallenge), or the AE does not recur (negative rechallenge).

An unexpected adverse drug event is any adverse drug event for which the specificity or severity is not consistent with the current IP.

#### 6.2.2.5 Seriousness of Adverse Events

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life threatening; this means that the patient was at risk of death at the time of the event; it does not mean that the event hypothetically might have caused death if it were more severe
- Requires hospitalization or prolongation in existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly or birth defect
- Is another important medical event (see below)

Important medical events that do not result in death, are not life threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they


may jeopardize the patient and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such events are:

- Intensive treatment in an emergency room or at home for allergic bronchospasm
- Blood dyscrasias or convulsions that do not result in inpatient hospitalization
- Development of drug dependency or drug abuse

Hospitalization for elective surgery or routine clinical procedures that are not the result of AE (eg, elective surgery for a pre-existing condition that has not worsened) need not be considered SAEs. If anything untoward is reported during the procedure, that occurrence must be reported as an AE, either 'serious' or 'nonserious' according to the usual criteria.

Suspected unexpected serious adverse reactions (SUSARs) are AEs that are associated with the use of the drug and are serious and unexpected.

### 6.2.2.6 Adverse Events of Special Interest

AEs of special interest in this study include the following:

- 1. Anaphylaxis and serious allergic reactions
- 2. Grades 2 to 5 injection site reaction, including erythema, pain, and induration (See APPENDIX 6)
- 3. Drug Induced Liver Injury (DILI) assessed following Hy's Law
- 4. Malignancy
- 5. Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, and disseminated tuberculosis
- 6. Cryptosporidiasis

## 6.2.2.6.1 Anaphylaxis and Serious Allergic Reactions

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria. <sup>42</sup> In the event of anaphylactic reaction or severe/serious hypersensitivity/allergic reaction, the patient must discontinue IP and emergency resuscitation measures implemented. In case of other mild to moderate hypersensitivity reaction, depending on the severity, the investigator may manage in accordance with the standard-of-care.

Anaphylaxis is highly likely when any one of the following 3 criteria is fulfilled:

- 1. Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (eg, generalized hives, pruritus, or flushing, swollen lips-tongue-uvula) and at least 1 of the following:
  - a. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow [PEF], hypoxemia)
  - b. Reduced blood pressure or associated symptoms of end-organ dysfunction (eg, hypotonia [collapse], syncope, incontinence)


- 2. Two or more of the following that occur rapidly after exposure to a likely allergen for that patient (minutes to several hours):
  - a. Involvement of the skin-mucosal tissue (eg, generalized hives, itch-flush, swollen lips-tongue-uvula)
  - b. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)
  - c. Reduced blood pressure or associated symptoms (eg, hypotonia [collapse], syncope, incontinence)
  - d. Persistent gastrointestinal symptoms (eg, crampy abdominal pain, vomiting)
- 3. Reduced blood pressure after exposure to known allergen for that patient (minutes to several hours):
  - a. Systolic blood pressure of less than 90 mm Hg or greater than 30% decrease from the patient's baseline

### **6.2.2.6.2 Injection Site Reactions**

Injection site reactions are to be captured and reported as AEs. These will include Grades 2 to 5 injection site erythema, pain, and induration (see APPENDIX 6), which are also captured as Adverse Events of Special Interest (See Section 6.2.2.6). The investigator should provide a clear description of the observed or reported AE including location and severity. All concomitant treatments used to treat injection site reactions should be recorded and captured in the eCRF, together with the AE of injection site reactions.

# 6.2.2.6.3 Potential Drug-Induced Liver Injury

Abnormal values in AST and/or ALT levels concurrent with abnormal elevations in total bilirubin level that meet the criteria outlined below in the absence of other causes of liver injury are considered potential cases of DILI, and as potential Hy's Law cases, and should always be considered important medical events. If symptoms compatible with DILI precede knowledge of serum chemical test abnormalities, liver enzyme measurements should be made immediately, regardless of when the next visit or monitoring interval is scheduled. In some cases, symptoms may be an early sign of injury and although typically less sensitive than serum enzyme elevations, they may indicate a need for prompt serum testing. An increase in liver enzymes should be confirmed by a repeated test within 48 to 72 hours following the initial test, prior to reporting of a potential DILI event. Patients will continue to have weekly or biweekly liver enzyme measurements until resolution or levels return to baseline.

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 6.2.2.7.2 for reporting details).

Potential DILI is defined as:

1. ALT or AST elevation  $> 3 \times ULN$ 

AND


2. Total bilirubin  $> 2 \times ULN$ , without initial findings of cholestasis (elevated serum alkaline phosphatase)

#### AND

3. No other immediately apparent possible causes of ALT or AST elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic

The patient should return to the investigational site and be evaluated as soon as possible, include laboratory tests, detailed history, and physical assessment. In addition to repeating measurements of AST and ALT, laboratory tests should include albumin, CK, total bilirubin, direct and indirect bilirubin, GGT, prothrombin time (PT)/International Normalized Ratio (INR), and alkaline phosphatase. A detailed history, including relevant information, such as review of ethanol, acetaminophen, recreational drug and supplement consumption, family history, occupational exposure, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and work exposure, should be collected. Further testing for acute hepatitis A, B, or C infection and liver imaging (eg, biliary tract) may be warranted. All cases confirmed on repeat testing as meeting the laboratory criteria defined above, with no other cause for liver function test (LFT) abnormalities identified at the time should be considered potential Hy's Law cases irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal LFTs. Such potential Hy's Law cases should be reported as SAEs.

Study drug discontinuation is considered if there is marked serum AST or ALT elevation or evidence of functional impairment (as indicated by rising bilirubin or INR, which represent substantial liver injury) that is related to study drug. Discontinuation of treatment should be considered if:

- ALT or AST > 8 × ULN
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks

Discontinuation of treatment must occur if:

- ALT or AST >3 × ULN and (total bilirubin > 2 × ULN or INR > 1.5)
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%)

### **6.2.2.6.4 Malignancy**

The identification of a malignancy event will be made by the study site and communicated to the sponsor or designee. AEs should be reported as serious per the criteria in Section 6.2.2.5.

After the first dose of study drug, when there is a decision to biopsy a potentially malignant tumor, lymph node, or other tissue, the investigator and/or consultant(s) should contact the sponsor clinicians or designee to discuss the issue and any decisions as soon as possible.


### 6.2.2.6.5 Specific Infections

Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, shingles, disseminated herpes simplex, or disseminated tuberculosis will be recorded as AEs of special interest.

Cryptosporidiosis is also considered an AE of special interest. Patients will be evaluated for cryptosporidium in the stool at screening, and as clinically indicated (eg, watery diarrhea) during the study. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

# 6.2.2.7 Reporting of Adverse Events

AE reporting will be carried out in accordance with applicable local regulations, including regulatory agency and IRB reporting requirements.

Each AE is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

### 6.2.2.7.1 Reporting of Pregnancy

As information is available, a pregnancy diagnosed during the study will be reported within 24 hours to the sponsor via the Pregnancy Notification and Outcome Form, including pregnancy in female patients who received study drug and female partners of male study patients who received study drug. The pregnancy should be followed to term and/or outcome and this outcome should also be reported to the sponsor via the Pregnancy Notification and Outcome Form. Pregnancy itself is not regarded as an AE or SAE unless there is complication.

In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an AE or SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live born, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as serious adverse events when the investigator assesses the neonatal death as related or possibly related to exposure to investigational product.


### 6.2.2.7.2 Reporting of Serious Adverse Events

The principal investigator is responsible for providing notification to the sponsor of any SAE via the Safety Adverse Event Form, whether deemed study drug related or not, that a patient experiences during their participation in this study within 24 hours of becoming aware of the event.

If an SAE is fatal or life threatening, notification to the sponsor must be made aware immediately, irrespective of the extent of available AE information. This timeframe also applies to additional new information (follow-up) on previously forwarded SAE reports as well as to the initial and follow-up reporting of exposure during pregnancy and exposure via breastfeeding cases. In the rare event that the investigator does not become aware of the occurrence of an SAE immediately (eg, if an outpatient study patient initially seeks treatment elsewhere), the investigator is to report the event within 24 hours after learning of it and document the time of his/her first awareness of the AE.

The principal investigator will review each SAE and evaluate the intensity and the causal relationship of the event to the study drug. All SAEs will be recorded from the time of first dose of study drug through the safety follow-up period (up to Day 270). SAEs occurring after the final follow-up visit and coming to the attention of the principal investigator must be reported only if there is (in the opinion of the principal investigator) reasonable causal relationship with the study drug.

As a minimum requirement, the initial notification should provide the following information:

- Study number
- Patient number
- Details of the SAE (verbatim details are sufficient for immediate notification)
- Criterion for classification as 'serious'
- Causality assessment (which may be updated in a follow-up report when sufficient information is available to make this classification)

Initial reports of SAEs must be followed later with detailed descriptions, including clear photocopies of other documents as necessary (eg, hospital reports, consultant reports, autopsy reports, etc), with the study patient's personal identifiers removed. All relevant information obtained by the principal investigator through review of these documents will be recorded and submitted to the sponsor within 24 hours of receipt of the information. If a new Safety Adverse Event Form is submitted, then the principal investigator must sign and date the form. The sponsor may also request additional information on the SAE, or clarification of omitted or discrepant information from the initial notification, which the principal investigator or an authorized delegate should submit to the sponsor within 24 hours of the request as possible.

#### **6.2.2.7.3** Reporting of Adverse Events of Special Interest

AEs of special interest will be reported to safety immediately or within 24 hours of the site becoming aware of the event and recorded as such on the Adverse Events eCRF and Safety Adverse Event Form


Potential DILI will be reported based on specifications mentioned in Section 6.2.2.6.3.

Each AE of special interest is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

### 6.2.2.8 Follow Up of Adverse Events

All AEs will be followed up through the safety follow-up visits. All SAEs experienced by a patient, irrespective of the suspected causality, will be monitored until the event has resolved, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the principal investigator and medical monitor, until there is a satisfactory explanation for the changes observed, or until the patient is lost to follow-up.

See Section 6.2.2.7.1 for details related to follow-up of pregnancy. See Section 6.2.2.6.3 for details related to follow-up of potential DILI. See Section 6.2.2.6.4 for details related to follow-up of malignancy.

#### 6.2.3 Vital Signs

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (Section 3.4). Vital signs will be assessed on Day 0 at predose and at Day 0, 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq 5$  minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection

#### 6.2.4 12-Lead Electrocardiograms

ECG will be assessed as specified in the Schedule of Assessments (Section 3.4). ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

The ECG will include all 12 standard leads and a Lead II rhythm strip on the bottom of the tracing. The ECG will be recorded at a paper speed of 25 mm/second. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QT interval corrected for heart rate using Fridericia's formula (QTcF).

All ECGs must be evaluated by a qualified physician or qualified designee for the presence of abnormalities and will be captured electronically and retained for future evaluation if required, up to the time of the clinical study report (CSR) completion.

#### 6.2.5 Physical Examinations

The full physical examination will be completed at screening and Day 0. It includes an assessment of general appearance and evaluation of head, eyes, ears, nose, mouth, throat, neck,


thyroid, lymph nodes, and extremities, and dermatologic, respiratory, cardiovascular, gastrointestinal, musculoskeletal, neurologic, and psychiatric systems.

The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Section 3.4). It includes evaluation of patient complaints and SLE disease-related issues, and will exclude the genitourinary system.

#### 6.2.6 C-SSRS

The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed by Columbia University researchers for the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening.<sup>43</sup>

The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Section 3.4). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

### **6.2.7** Injection Site Reactions

Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (Section 3.4). Local injection site reactions will be assessed at 2 hours postdose at baseline, and predose for each injection after baseline. Injection site reactions should be managed according to the standard of care. Injection site reactions, Grades 2 to 5, are to be reported as AEs of special interest (see Section 6.2.2.7.3).

#### 6.2.8 Immunogenicity

The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (Section 3.4). Blood samples (4 mL) to provide approximately 1.5 mL of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K<sub>2</sub>EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only analyzed by a central lab if the patient had a positive ADA on Day 90.

After the first dose, if a patient tests positive in the validated confirmatory ADA assay, a sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay by a central lab.


# **6.3** Efficacy Assessments

All efficacy assessments will be performed at times defined in the Schedule of Assessments (Section 3.4).

#### **6.3.1 SLEDAI-2K**

The SLEDAI-2K is a validated instrument that measures disease activity in SLE patients at the time of the visit and in the previous 30 days. It is a global index and includes 24 clinical and laboratory variables that are weighted by the type of manifestation, but not by severity. The total score falls between 0 and 105, with higher scores representing increased disease activity. The SLEDAI-2K has been shown to be a valid and reliable disease activity measure in multiple patient groups. A SLEDAI -2K of 6 or more generally represents moderately to severely active disease. 44

#### 6.3.2 BILAG 2004

The BILAG-2004 index is an organ-specific 97-question assessment based on the principle of the doctor's intent to treat. Only clinical features attributable to SLE disease activity are to be recorded and based on the patient's condition in the last 4 weeks compared with the previous 4 weeks. It will be scored as not present (0), improved (1), the same (2), worse (3), or new (4). Disease activity is graded separately for 9 body systems to 5 different grades (A to E) as follows: A ("Active") is very active disease, B ("Beware") is moderate activity, C ("Contentment") is mild stable disease, D ("Discount") is inactive now but previously active, and E ("Excluded") indicates the organ was never involved. A shift from BILAG-2004 Grade A or B to a lower grade indicates a clinically relevant change in disease activity as the BILAG-2004 grades mirror the decision points for treatment interventions.

Only investigators that complete BILAG-2004 training will be allowed to perform the BILAG-2004 assessments. Preferably, the same investigator should evaluate the patient at each BILAG-2004 assessment from screening to study completion. The investigator must maintain documentation with descriptive details supporting the BILAG-2004 scoring (eg, chart, worksheet, clinic notes, and labs) at each visit.

See APPENDIX 5 for detailed specifications.

#### 6.3.3 PGA of Disease Activity

The PGA is used to assess investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients". PGA worsening is defined as an increase of  $\geq$  30 mm from baseline.

When scoring the PGA, the assessor should always look back at the score from the previous visit.


# 6.3.4 Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response

#### 6.3.4.1 SRI-4 Response

The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. Response based on the SRI-4 is defined by:

1)  $\geq$  4-point reduction in SLEDAI-2K global score, 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B), and 3) no deterioration from baseline in the PGA by  $\geq$  30 mm. The SRI-4 response in patients with moderate to severe SLE is associated with broad improvements in clinical and patient-reported outcomes. <sup>45</sup>

### 6.3.4.2 SRI-5 and SRI-6 Response

Like the SRI-4, the SRI-5 and SRI-6 are composite indices of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. However, the SRI-5 and SRI-6 are computed with a minimal five-point or six-point improvement in SLEDAI-2K being required, respectively. 46

### 6.3.4.3 BICLA Response

The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and PGA. BICLA response is defined as 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (eg, all B [moderate disease] scores falling to C [mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4)  $\leq$  10% deterioration in PGA score and 5) no treatment failure.<sup>44</sup> It is driven primarily by the BILAG, and has been used in Phase 2 and 3 mAb studies.<sup>47</sup>

For the endpoints of BICLA response at Days 210, 240, and 270, patient scores will be completed and response determined.

### 6.3.5 CLASI Response

The CLASI is a comprehensive tool for assessment of disease activity and damage in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity. <sup>48</sup> Response is defined as 50% improvement from baseline in "A" or "B" scores. This assessment will be applied to all patients as all are required to have cutaneous disease activity.

For the secondary efficacy endpoint of CLASI response at Day 210, patient scores on MAD and POC studies will be compared with baseline for 50% improvement.

#### 6.3.6 ACR-28 Joint Count

The ACR-28 joint count will evaluate the number of tender and swollen joints in the shoulder, elbow, wrist, hand, knee joints. Joints of the feet are excluded.


#### 6.4 Other Variables

#### 6.4.1 SLICC/ACR Damage Index

The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in patients with SLE regardless of cause, with demonstrated content, face, criterion, and discriminant validity. It will be performed on Days 0 and 180.

#### 6.4.2 **PROs**

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the CCI and the CCI and will be assessed as specified in the Schedule of Assessments (Section 3.4).



#### 6.5 Pharmacokinetic Assessments

During the MAD Phase 1b (all sites) and POC Phase 2 (select sites only) parts of the study, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to Table 1 and Table 2.

Plasma concentrations of BOS161721 will be measured using a validated immunoassay. The PK parameters will be calculated from the plasma concentration actual time profiles.

## 6.6 Pharmacodynamic Assessments

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (Section 3.4) for each of the following parameters:

• pSTAT3 (predose [trough] samples only Phase 1b)

• Antibodies: CC

• Plasma complement (CCI)

• Plasma CCI and CCI

• Whole blood for leukocyte immunophenotype


# 6.7 Pharmacokinetic/Pharmacodynamic Relationship

Evidence of any PK/PD relationships will be evaluated between BOS161721 plasma concentrations and the available PD endpoints and biomarkers.

#### **6.8** Protocol Deviations

Protocol deviations will be documented during the study.

#### 7 STUDY DRUG MANAGEMENT

# 7.1 Description

#### 7.1.1 Formulation



Additional information regarding dose preparation will be provided in a separate Pharmacy Manual.

### 7.1.2 Storage

All supplies of BOS161721 or placebo must be stored in accordance with the manufacturer's instructions. BOS161721 or placebo will be stored in a securely locked area, accessible to authorized persons only, until needed for dosing.

Information regarding storage and dose preparation will be provided in a separate Pharmacy Manual.

# 7.2 Packaging and Shipment

Investigational medicinal products will be supplied by Boston Pharmaceuticals, Inc. Investigational medicinal products will be packaged and labeled according to applicable local and regulatory requirements.

#### 7.3 Dose and Administration

Details of dosing are provided in Section 3.1.

Each unit dose will be prepared by a qualified staff member. The vials of investigational product (IP) will appear identical and will have a "blinded" label on the vials that will state mg or placebo. When the site goes into the IWRS to request the patient kit(s), the IWRS will assign the


BOS161721 Boston Pharmaceuticals, Inc.


appropriate number of kits (regardless of assignment to placebo or active treatment) per the dose (ie, CCI). If a patient is randomized to the placebo arm, they will receive the matching number of kits.

The designated staff member (or designee under the direction of the designated staff member) will dispense BOS161721 or placebo for each patient according to the protocol, randomization list, and Pharmacy Manual, if applicable.

After receiving sponsor approval in writing, the investigational site is responsible for returning all unused or partially used BOS161721 or placebo to the sponsor or designated third party or for preparing BOS161721 or placebo for destruction via incineration.

Further details are found in a separate Pharmacy Manual.

# 7.4 Accountability

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Products returned to the pharmacy will be stored under the same conditions as products not yet dispensed. The returned products should be marked as 'returned' and kept separate from the products not yet dispensed.

All dispensing and accountability records will be available for sponsor review after database lock procedures are completed. During safety monitoring, the drug accountability log will be reconciled with the products stored in the pharmacy.

# 7.5 Prohibited Concomitant Therapy

Prohibited concomitant medications are discussed in Section 4.6 and APPENDIX 4 and will be listed as protocol violations if taken when not permitted.

# 7.6 Compliance

Dosing will be performed by trained, qualified personnel designated by the principal investigator. The date and time of dosing will be documented on each dosing day. Comments will be recorded if there are any deviations from the planned dosing procedures.

#### 8 STATISTICS

The following analyses are planned:

- An IA will be performed during the last cohort of the MAD portion to determine dose selection for the POC part of the study.
- The final analysis will be performed when all patients have completed the POC safety follow-up or withdrawn from the study.
- Safety analyses will be performed for DMC reviews throughout the study to evaluate dose escalation decisions and accumulating safety data. The frequency and details of the


content and format of the safety review meetings will be described in the SAP and/or DMC charter.

All statistical analyses will be performed using Statistical Analysis Software (SAS®) Version 9 or higher.

The following standards will be applied for the analysis unless otherwise specified. Data will be summarized descriptively by treatment and overall for each study portion. For the MAD part of the study, BOS161721 will be summarized overall and by each dose level, and placebo patients from each cohort will be combined. Select parameters may be summarized using patients from both study parts. Statistical testing will be performed on data from the Phase 2 portion only.

Continuous data will be summarized using number, mean, standard deviation (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, median, and maximum. Categorical data will be summarized by treatment group using frequency tables (number and percentage). Time to event data will be summarized using counts, medians, 25<sup>th</sup> and 75<sup>th</sup> percentiles, and standard error. All data will be listed for all patients.

Statistical inference will be based on a 2-tailed test with an overall 0.10 level of significance, unless stated otherwise

The effects of noncompliance, background therapy use, treatment discontinuations, premature withdrawal from study and covariates will be assessed to determine the impact on the general applicability of results from this study. Exploratory analyses of the data will be conducted as deemed appropriate. Any deviations from the planned analyses will be described and justified in the final integrated CSR.

Protocol deviations and prohibited medications that define medication failures will be fully assigned and documented before database lock and unblinding.

Further details of the analysis, including the handling of missing data, transformations and other data handling procedures will be provided in the SAP.

# 8.1 Sample Size

Sample size in the Phase 1b part of the study is based on operational consideration.

The sample size in the Phase 2 portion is based on the primary endpoint, SRI-4 Response at Day 210. Approximately 156 additional patients will be randomized in a 2:1 ratio to BOS161721 versus placebo to achieve 132 evaluable patients in the FAS. This assumes 24 patients will drop prior to having received treatment and an evaluable post-baseline efficacy measure. Enrollment and randomization will be monitored in a blinded fashion and increased if needed to ensure at least 132 patients are randomized into the FAS.

A total of 132 patients randomized provides more than 80% power to detect a treatment difference of 25% in SRI-4 response rates at Day 210, based on a targeted 2-sided significance level of 10% and using a 2-sided Pearson's chi-squared test. This assumes of a response rate of 65% for BOS161721 and 40% for placebo, where missing data at Day 210 is carried forward


from most recent non-missing result and patients are treated as a non-responder if a prohibited medication defined as a medication failure occurs.

#### **8.2** Statistical Methods

#### 8.2.1 Analysis Populations

The primary efficacy analysis will be based on the FAS, defined as all patients who receive at least 1 dose of study treatment and at have least 1 evaluable post-baseline efficacy evaluation. FAS analyses will be conducted on the basis of the randomized treatment.

A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be identified based on blinded data prior to study unblinding. PP analyses will be conducted on the basis of the randomized treatment.

Safety analyses will be based on the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. Safety analyses will be conducted on the basis of actual treatment received.

Pharmacokinetic analysis will be conducted on the PK analysis set, defined as the FAS with sufficient concentration data for the calculation of PK parameters.

#### 8.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized using all randomized patients.

#### 8.2.3 Primary Efficacy Endpoint(s)

The proportion of patients who achieve a SRI-4 response at Day 210 will be assessed via Pearson's chi-squared analysis. The primary efficacy endpoint will be analyzed using the FAS and if needed repeated in the PP analysis set. Missing values will be addressed by employing a last observation carried forward (LOCF) analysis. Other imputation methods may be employed as a sensitivity analysis and will be described in the SAP. Additional analyses exploring impact of baseline factors such as baseline disease severity, race, and other characteristics may be performed.

Patients that received prohibited medications or unallowable CS usage as described in Section 4.6 will be considered "medication failures" and will be treated as non-responders for the primary efficacy analysis. Patients that received an allowable CS burst but having missing data at Day 210 will considered a medication failure and will be treated as non-responders for the primary efficacy analysis. The determination of medication failures will be reviewed using blinded data and finalized prior to unblinding.

The superiority of BOS161721 relative to placebo will be evaluated. If the proportion of SRI-4 responders for the selected POC dose in BOS161721 arm is higher than that of the placebo arm, then BOS161721 will be considered superior to placebo if the 2-sided p-value is less than 0.10.


Secondary and exploratory endpoints for this POC portion will be evaluated based on the same statistical hypothesis.

#### 8.2.4 Secondary Efficacy Endpoint(s)

Binary efficacy endpoints will be assessed via Pearson's chi-squared analysis. Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) and treatment will be compared using the F-test. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test. The secondary efficacy endpoints will be analyzed on the FAS and if needed repeated in the PP analysis set. Details including handling of missing data and "medication failures" will be available in the SAP.

#### 8.2.5 Analysis of Safety

### 8.2.5.1 Safety Analysis

Safety analyses will be performed on the SS. AE data will be coded to system organ class and preferred term using MedDRA. The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term, will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be coded using the WHO Drug dictionary. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters will be summarized at each individual visit.

#### 8.2.6 Pharmacokinetic and Pharmacodynamic Data

# 8.2.6.1 Analysis of Pharmacokinetic Data

PK parameters will be calculated from concentration data collected during the MAD Phase 1b portion of the study using non-compartmental analysis and include the following:

• Cmax, Tmax, AUC, t1/2, CL, Vd

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:

- A listing of all plasma BOS161721 concentrations by patient at actual times post dose;
- A descriptive summary of plasma BOS161721 concentrations. Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.


#### 8.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Exploratory analyses examining the relationship between PD parameters and PK concentration and PK parameters will be performed.

#### 8.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints.

# 8.3 Interim Analysis and Power

One IA is planned for this study and will be conducted at the time of the POC decision for dose selection.

Since there is no IA during the POC part of the study, there is no impact on the type 1 error.

#### 9 ETHICS AND RESPONSIBILITIES

#### 9.1 Good Clinical Practice

The procedures set out in this protocol are designed to ensure that the sponsor and the principal investigator abide by the principles of the International Council for Harmonisation (ICH) guidelines on GCP and the Declaration of Helsinki (Version 2013). The clinical study also will be carried out in the keeping with national and local legal requirements (in accordance with US IND regulations [21 CFR 56]).

#### 9.2 **DMC**

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for BOS161721. The recommendations made by the DMC (ie, dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.

The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the


accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) suggest dose for POC portion of the study as described in Section 3.1.1.3.

The DMC considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

The DMC will have access to unblinded treatment information during the clinical trial. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of BOS161721 treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.

# 9.3 Institutional Review Board/Independent Ethics Committee

Independent Ethics Committees (IEC)/Institutional Review Boards (IRB) must meet the guidelines set out by the U.S. Food and Drug Administration (FDA) and conform to local laws and customs where appropriate. Written IRB/IEC approval for the protocol and the signed ICF must be obtained and transmitted to Boston Pharmaceuticals or representative before the study can be initiated. The IRB/IEC must be informed of and approve all protocol amendments. The investigator will ensure that this study is conducted in full conformance with all applicable local and regional laws and regulations. The complete text of the World Medical Association Declaration of Helsinki is given in APPENDIX 2.

#### 9.4 Informed Consent

Before each patient undergoes any protocol required assessments or procedure, the written informed consent will be obtained according to the regulatory and legal requirements of the participating country. As part of this procedure, the principal investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study patient should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The principal investigator or designee will provide the sponsor with a copy of the IRB-approved ICF prior to the start of the study.

The informed consent document must be signed and dated; 1 copy will be handed to the patient and the principal investigator will retain a copy as part of the clinical study records. The principal investigator will not undertake any investigation specifically required for the clinical study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented.


If the informed consent document is revised, it must be reviewed and approved by the responsible IRB/IEC. Patients currently enrolled may need to sign this revision (based on IRB/IEC requirements) and all future patients enrolled in the clinical study will be required to sign this revised ICF.

### 9.5 Records Management

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes. The principal investigator or designee will cooperate with the sponsor's representative(s) for the periodic review of study documents to ensure the accuracy and completeness of the data capture system at each scheduled monitoring visit.

Electronic consistency checks and manual review will be used to identify any errors or inconsistencies in the data. This information will be provided to the respective study sites by means of electronic or manual queries.

The principal investigator or designee will prepare and maintain adequate and accurate study documents (medical records, ECGs, AE and concomitant medication reporting, raw data collection forms, etc.) designed to record all observations and other pertinent data for each patient receiving BOS161721 or placebo.

The principal investigator will allow sponsor representatives, contract designees, authorized regulatory authority inspectors, and the IRB to have direct access to all documents pertaining to the study.

Electronic case report forms are required and should be completed for each randomized patient. It is the principal investigator's responsibility to ensure the accuracy, completeness, legibility, and timeliness of the data reported on the patients' eCRF. Electronic case report forms should be completed in a timely fashion to support the study timelines. Source documentation supporting the eCRF data should indicate the patient's participation in the study and should document the dates and details of study procedures, AEs, and patient status. The principal investigator or designated representative should complete and the principal investigator should verify the source documents as the information is collected. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the Sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes.

#### 9.6 Source Documentation

The documents that will form the source data for the clinical study (eg, patient charts, laboratory reports) must be defined and documented in the in-house study master file prior to the start of the study. Data on the eCRFs which will be checked against source data during monitoring visits


must also be defined and documented in the in-house study master file including the percentage of each of the source data to be verified and the percentage of patients' eCRFs to be monitored.

# 9.7 Study Files and Record Retention

According to ICH guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of BOS161721. However, these documents should be retained for a longer period if required by the applicable legal requirements.

#### 10 AUDITING AND MONITORING

Throughout the course of the study, the study monitor will make frequent contacts with the investigator. This will include telephone calls and on-site visits. The study will be routinely monitored to ensure compliance with the study protocol and the overall quality of data collected. During the on-site visits, the eCRFs will be reviewed for completeness and adherence to the protocol. As part of the data audit, source documents will be made available for review by the study monitor. The study monitor may periodically request review of the investigator study file to assure the completeness of documentation in all respects of clinical study conduct. The study monitor will verify that each patient has proper consent documentation from the patient and/or patient's authorized representative for study procedures and for the release of medical records to the sponsor, FDA, other regulatory authorities, and the IRB. The study monitor will also verify that assent was obtained for patients not capable of providing informed consent or that documentation is provided by the investigator explaining why the patient was unable to provide assent. The investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the investigator will permit inspection of the study files by authorized representatives of the regulatory agencies. On completion of the study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

Throughout the course of the study, the medical monitor will determine eligibility of all screened patients, will address any medical issues that might arise, clarify medical questions, review patient safety data (eg, AE/SAE, laboratory, and ECG), and partner with the study team in the overall study management. The study medical monitoring plan will document additional details of the study medical oversight and monitoring.

#### 11 AMENDMENTS

Protocol modifications, except those intended to reduce immediate risk to study patients, may be made only by Boston Pharmaceuticals. A protocol change intended to eliminate an apparent immediate hazard to patients may be implemented immediately, provided the IRB/IEC is notified within 5 days.

Any permanent change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB/IEC and the investigator must await approval before


implementing the changes. Boston Pharmaceuticals will submit protocol amendments to the appropriate regulatory authorities for approval.

If in the judgment of the IRB/IEC, the investigator, and/or Boston Pharmaceuticals, the amendment to the protocol substantially changes the study design and/or increases the potential risk to the patient and/or has an impact on the patient's involvement as a study participant, the currently approved written ICF will require similar modification. In such cases, informed consent will be renewed for patients enrolled in the study before continued participation.

#### 12 STUDY REPORT AND PUBLICATIONS

Boston Pharmaceuticals is responsible for preparing and providing the appropriate regulatory authorities with clinical study reports according to the applicable regulatory requirements.

By signing the protocol, the principal investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the principal investigator's name, address, qualifications, and extent of involvement.

The principal investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted and obtained approval from the sponsor in advance.

#### 13 STUDY DISCONTINUATION

Both Boston Pharmaceuticals and the principal investigator reserve the right to terminate the study at the investigator's site at any time. Should this be necessary, Boston Pharmaceuticals or a specified designee will inform the appropriate regulatory authorities of the termination of the study and the reasons for its termination, and the principal investigator will inform the IRB/IEC of the same. In terminating the study Boston Pharmaceuticals and the principal investigator will assure that adequate consideration is given to the protection of the patients' interests.

#### 14 CONFIDENTIALITY

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from Boston Pharmaceuticals, except to the extent necessary to obtain informed consent from patients who wish to participate in the trial or to comply with regulatory requirements. However, authorized regulatory officials, IRB/IEC personnel, Boston Pharmaceuticals, and its authorized representatives are allowed full access to the records.

Identification of patients and eCRFs shall be by initials, birthdate, or patient number. Documents that identify the patient (eg, the signed informed consent document) must be maintained in confidence by the principal investigator. If required, the patient's full name may be made known to an authorized regulatory agency or other authorized official.


### 15 REFERENCES

1 Urowitz MB, Gladman DD. How to improve morbidity and mortality in systemic lupus erythematosus. Rheumatology 2000;39:238-44.

- 2 Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, et al. Morbidity and Mortality in Systemic Lupus Erythematosus During a 10-Year Period. Medicine 2003;82(5):299-308.
- 3 Pons-Estel GJ, Alarcón GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010;39(4):257. Epub 2009 Jan 10.
- 4 Kanta H, Mohan C. Three Checkpoints in lupus development: central tolerance in adaptive immunity, peripheral amplification by innate immunity, and end-organ inflammation. Genes and Immunity 2009;10:390-6.
- 5 Dall'Aqua WF, Kiener PA, Wu H. Properties of Human IgG1s Engineered for Enhanced Binding to the Neonatal Fc Receptor (FcRn). J Biol Chem. 2006 Aug 18, 281(33):23514-24.
- 6 Spolski R, Leonard WJ. The Yin and Yang of interleukin-21 in allergy, autoimmunity and cancer. Curr Opin Immunol. 2008a;20:295-301.
- 7 Asao H, Okuyama C, Kumaki S, Ishii N, Tsuchiya S, Foster D, et al. Cutting edge: the common gamma-chain is an indispensable subunit of the IL-21 receptor complex. J Immunol. 2001;167:1-5.
- 8 Habib T, Senadheera S, Weinberg K, Kaushansky K. The common gamma chain (gamma c) is a required signaling component of the IL-21 receptor and supports IL-21-induced cell proliferation via JAK3. Biochemistry. 2002;41:8725-31.
- 9 Spolski R, Leonard WJ. Interleukin-21: basic biology and implications for cancer and autoimmunity. Annu Rev Immunol. 2008b;26:57-79.
- 10 Puga I, Cols M, Barra CM, He B, Cassis L, Gentile M, et al. B-cell-helper neutrophils stimulate the diversification and production of immunoglobulin in the marginal zone of the spleen. Nat Immunol. 2011;13(2):170-80.
- 11 Costanzo A, Chimenti MS, Botti E, Caruso R, Sarra M, Monteleone G. IL-21 in the pathogenesis and treatment of skin diseases. J Dermatol Sci. 2010;60(2):61-6.
- 12 Avery DT, Bryant VL, Ma CS, de Waal Malefy R, Tangye SG. IL-21-induced isotype switching to IgG and IgA by human naive B cells is differentially regulated by IL-4. J Immunol. 2008;181:1767-79.
- 13 Rasmussen TK, Andersen T, Bak, RO, Yiu G, Sorensen CM, Stengaard-Pedersen K, et al. Overexpression of microRNA-155 increases IL-21 mediated STAT3 signaling and IL-21 production in systemic lupus erythematosus. Arthritis Research & Therapy 2015;17(154)


- 14 Ettinger R, Kuchen S, Lipsky PE. The role of IL-21 in regulating B-cell function in health and disease. Immunol Rev. 2008;223:60-86.
- 15 Caprioli F, Sarra M, Caruso R, Stolfi C, Fina D, Sica G, et al. Autocrine regulation of IL-21 production in human T lymphocytes. J Immunol. 2008;180(3):1800-7.
- 16 Yang L, Anderson DE, Baecher-Allan C, Hastings WD, Bettelli E, Oukka M, et al. IL-21 and TGF-beta are required for differentiation of human T(H)17 cells. Nature. 2008;454(7202):350-2.
- 17 Tangye SG, Ma CS, Brink R, Deenick EK. The good, the bad and the ugly TFH cells in human health and disease. Nat Rev Immunol. 2013;13(6):412-26.
- 18 Fantini MC, Rizzo A, Fina D, Caruso R, Becker C, Neurath MF, et al. IL-21 regulates experimental colitis by modulating the balance between Treg and Th17 cells. Eur J Immunol. 2007;37(11):3155-63.
- 19 Peluso I, Fantini MC, Fina D, Caruso R, Boirivant M, MacDonald TT, et al. IL-21 counteracts the regulatory T-cell-mediated suppression of human CD4+ T lymphocytes. J Immunol. 2007;178(2):732-9.
- 20 Hippen KL, Bucher C, Schirm DK, Bearl AM, Brender T, Mink KA, et al. Blocking IL-21 signaling ameliorates xenogeneic GVHD induced by human lymphocytes. Blood. 2012;119(2):619-28.
- 21 Davis ID, Skrumsager BK, Cebon J, Nicholaou T, Barlow JW, Moller NP, et al. An open-label, two-arm, phase I trial of recombinant human interleukin-21 in patients with metastatic melanoma. Clin Cancer Res. 2007;13:3630-6.
- 22 Frederiksen KS, Lundsgaard D, Freeman JA, Hughes SD, Holm TL, Skrumsager BK, et al. IL-21 induces in vivo immune activation of NK cells and CD8(+) T-cells in patients with metastatic melanoma and renal cell carcinoma. Cancer Immunol Immunother. 2008;57(10):1439-49.
- 23 Karrich JJ, Jachimowski LC, Nagasawa M, Kamp A, Balzarolo M, Wolkers MC, et al. IL-21- stimulated human plasmacytoid dendritic cells secrete granzyme B, which impairs their capacity to induce T-cell proliferation. Blood. 2013;121(16):3103-11.
- 24 Lindner S, Dahlke K, Sontheimer K, Hagn M, Kaltenmeier C, Barth TF, et al. Interleukin-21-induced granzyme B-expressing B-cells infiltrate tumors and regulate T-cells. Cancer Res. 2013;73(8):2468-79.
- 25 Monteleone G, Caruso R, Fina D, Peluso I, Gioia V, Stolfi C, et al. Control of matrix metalloproteinase production in human intestinal fibroblasts by interleukin 21. Gut. 2006;55(12):1774-80.
- 26 Nakou M, Papadimitraki ED, Fanouriakis A, Bertsias GK, Choulaki C, Goulidaki N, et al. Interleukin-21 is increased in active systemic lupus erythematosus patients and contributes to the generation of plasma B-cells. Clin Exp Rheumatol. 2013;31(2):172-9.


- 27 Li Q, Liu Z, Dang E, Jin L, He Z, Yang L, et al. Follicular helper T-cells (Tfh) and IL-21 involvement in the pathogenesis of bullous pemphigoid. PLoS One. 2013;8(7):e68145.
- 28 Liu R, Wu Q, Su D, Che N, Chen H, Geng L, et al. A regulatory effect of IL-21 on T follicular helper-like cell and B-cell in rheumatoid arthritis. Arthritis Res Ther. 2012;14(6):R255.
- 29 Kang KY, Kim HO, Kwok SK, Ju JH, Park KS, Sun DI, et al. Impact of interleukin-21 in the pathogenesis of primary Sjögren's syndrome: increased serum levels of interleukin-21 and its expression in the labial salivary glands. Arthritis Res Ther. 2011;13(5):R179.
- 30 Terrier B, Geri G, Chaara W, Allenbach Y, Rosenzwajg M, Costedoat-Chalumeau N, et al. Interleukin-21 modulates Th1 and Th17 responses in gianT-cell arteritis. Arthritis Rheum. 2012a;64(6):2001-11.
- 31 Terrier B, Costedoat-Chalumeau N, Garrido M, Geri G, Rosenzwajg M, Musset L, et al. Interleukin 21 correlates with T-cell and B-cell subset alterations in systemic lupus erythematosus. J Rheumatol. 2012b;39(9):1819-28.
- 32 International Conference on Harmonisation. Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals S6 (R1). 2011.
- 33 Wang W, Wang EQ, Balthasar JP. Monoclonal Antibody Pharmacokinetics and Pharmacodynamics. Clin Pharm & Ther 2008; 84(5):548-58.
- 34 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 35 Elsaesser H, Sauer K, Brooks DG. IL-21 is required to control chronic viral infection. Science. 2009;324(5934):1569-72
- 36 Kotlarz D, Zietara N, Uzel G, Weidemann T, Braun CJ, Diestelhorst J, et al. Loss-of-function mutations in the IL-21 receptor gene cause a primary immunodeficiency syndrome. J Exp Med. 2013;210(3):433-43.
- 37 Hunter PR, Nichols G. Epidemiology and clinical features of Cryptosporidium infection in immunocompromised patients. Clinical microbiology reviews. 2002;15(1):145-54.
- 38 Desjardins M, Mazer BD. B-cell memory and primary immune deficiencies: interleukin-21 related defects. Curr Opin Allergy Clin Immunol. 2013;13(6):639-45.
- 39 Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. *Nephron*. 1976;16(1):31-41.


- 40 Guidelines for Using the QuantiFERON®-TB Gold Test for Detecting Mycobacterium tuberculosis Infection, US: http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5415a4.htm.
- 41 NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, available at https://evs.nci.nih.gov/ftp1/CTCAE/About.html.
- 42 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 43 Posner K, Melvin G a, Stanley B, Oquendo M a, Gould M. Factors in the assessment of suicidality in youth. *CNS Spectr*. 2007;12(2):156-162.
- 44 Castrejon I, Tani C, Jolly M, Huang A, Mosca M. Indices to assess patients with systemic lupus erythematosus in clinical trials, long-term observational studies, and clinical care. Clin Exp Rheumatol 2014; 32(85):S85-95.
- 45 Furie R, Wang L, Drappa J, Illei G. Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] Response Is Associated with Global Benefit in Patients with Moderate to Severe SLE [abstract]. *Arthritis Rheumatol.* 2016; 68 (suppl 10).
- 46 Thanou A, Chakravarty E, James JA, Merrill JT. Which outcome measures in SLE clinical trials best reflect medical judgment? Lupus Science & Medicine 2014;1:e000005. doi:10.1136/lupus-2013-000005.
- 47 Wallace DJ, Kalunian K, Petri MA, Strand V, Houssiau FA, Pike M, et al. Efficacy and safety of epratuzumab in patients with moderate/severe active systemic lupus erythematosus: results from EMBLEM, a phase IIb, randomised, double-blind, placebo-controlled, multicentre study. *Ann Rheum Dis* 2014;73:183-90.
- 48 Albrecht J, Taylor L, Berlin JA, Dulay S, Ang G, Fakharzadeh S. The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index): An Outcome Instrument for Cutaneous Lupus Erythematosus. J Invest Derm. 2005;125(5):889-94.
- 49 Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is Valid, and Renal and Pulmonary Organ Scores are Predictors of Sever Outcome in Patients with Systemic Lupus Erythematosus. Br J Rheumatol. 1996;35:248-54.

50 **CCI** 


# 16 APPENDICES

# APPENDIX 1 NAMES OF STUDY PERSONNEL




### APPENDIX 2 DECLARATION OF HELSINKI

#### WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI

Ethical Principles
For
Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly
Helsinki, Finland, June 1964
and amended by the
29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
and the

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### A. INTRODUCTION

The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.

It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.

The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my subject will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the subject's interest when providing medical care which might have the effect of weakening the physical and mental condition of the subject."

Medical progress is based on research, which ultimately must rest in part on experimentation involving human subjects.

In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.

The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic, and therapeutic procedures and the understanding of the etiology and pathogenesis of disease. Even the best-proven prophylactic, diagnostic, and therapeutic methods must continuously be challenged through research for their effectiveness, efficiency, accessibility, and quality.


In current medical practice and in medical research, most prophylactic, diagnostic, and therapeutic procedures involve risks and burdens.

Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.

Research investigators should be aware of the ethical, legal, and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal, or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### B. BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.

Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.

Appropriate caution must be exercised in the conduct of research, which may affect the environment, and the welfare of animals used for research must be respected.

The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any SAEs. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.

The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles enunciated in this Declaration.

Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a subject of the research, even though the subject has given consent.

Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the


subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.

Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.

Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.

Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.

The subjects must be volunteers and informed participants in the research project.

The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the subject's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.

In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.

When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.

For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the investigator must obtain informed consent from the legally authorized representative in accordance with applicable law. These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.

When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the investigator must obtain that assent in addition to the consent of the legally authorized representative.

Research on individuals from whom it is not possible to obtain consent, including proxy or advance consent, should be done only if the physical/mental condition that prevents obtaining


informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.

Both authors and publishers have ethical obligations. In publication of the results of research, the investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic, or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the subjects who are research subjects.

The benefits, risks, burdens, and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic, or therapeutic method exists.

At the conclusion of the study, every subject entered into the study should be assured of access to the best-proven prophylactic, diagnostic, and therapeutic methods identified by the study.

The physician should fully inform the subject which aspects of the care are related to the research. The refusal of a subject to participate in a study must never interfere with the subject-physician relationship.

In the treatment of a subject, where proven prophylactic, diagnostic, and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the subject, must be free to use unproven or new prophylactic, diagnostic, and therapeutic measures, if in the physician's judgment it offers hope of saving life, re-establishing health, or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases, new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.


# APPENDIX 3 COMMONLY USED CORTICOSTEROID EQUIVALENTS

| Medication | Dose Equivalence |
|--------------------|------------------|
| Prednisone | 20 mg |
| Cortisone | 100 mg |
| Hydrocortisone | 80 mg |
| Prednisolone | 20 mg |
| Methylprednisolone | 16 mg |
| Triamcinolone | 16 mg |
| Budesonide | 4 mg |
| Dexamethasone | 3 mg |
| Bethamethasone | 2.4 mg |


# APPENDIX 4 MEDICATION WASHOUT PERIODS

# WASHOUT TIMES OF MEDICATIONS BASED ON 5 HALF-LIVES

| Medication | Discontinuing Prior to Signing Consent |
|---|---|
| Abatacept (CTLA4Ig) | 24 weeks |
| Alefacept | 12 weeks |
| AMG 623 (blisibimod) | 24 weeks |
| Anifrolumab | 12 weeks |
| Atacicept (TACI-Ig) | 12 weeks |
| Belimumab | 24 weeks |
| Cyclophosphamide | 24 weeks |
| Cyclosporine (except for CSA eye drops) | 4 weeks for oral and 8 weeks for topical |
| Danazol | 4 weeks |
| Dapsone | 4 weeks |
| Eculizumab | 12 weeks |
| Efalizumab | 12 weeks |
| Epratuzumab | 24 weeks |
| Intravenous globulin | 4 weeks |
| Leflunomide | 8 weeks (4 weeks for washout with |
| | cholestyramine) |
| Lenalidomide with cholestiramine | 8 weeks |
| Lupuzor | 12 weeks |
| Memantine | 4 weeks |
| Natalizumab | 24 weeks |
| Ocrelizumab | 48 weeks (or 24 weeks with recovery of B cell) |
| Pimecrolimus | 4 weeks |
| Plasmapheresis | 24 weeks |
| Retinoids (oral or topical) | 4 weeks |
| Rituximab | 48 weeks (or 24 weeks with recovery of B cell) |
| Sirolimus | 4 weeks |
| Tacrolimus | 4 weeks |
| Thalidomide | 8 weeks |
| Tocilizumab | 12 weeks |


# APPENDIX 5 BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA)




# APPENDIX 6 INJECTION SITE REACTION GRADING SCALE

| Adverse event<br>Injection site reaction | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade<br>5 |
|---|---|---|---|---|---|
| Definition: A disorder<br>characterized by an<br>intense adverse reaction<br>(usually immunologic)<br>developing at the site of<br>an injection | Tenderness with<br>or without<br>associated<br>symptoms (eg,<br>warmth,<br>erythema,<br>itching) | Pain;<br>Lipodystrophy;<br>Edema;<br>phlebitis | Ulceration or<br>necrosis;<br>Severe tissue<br>damage;<br>Operative<br>intervention<br>indicated | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>indicated | Death |
| Pain | Mild pain | Moderate pain;<br>limiting<br>instrumental ADL | Severe pain;<br>limiting self-<br>care ADL | - | - |
| Rash<br>maculopapular/Erythema<br>/Induration | Macules/papules<br>covering <10%<br>BSA with or<br>without | Macules/papules<br>covering 10% -<br>30% BSA with or<br>without symptoms | Macules/papul<br>es covering<br>> 30% BSA<br>with or | - | - |
| Definition: A disorder<br>characterized by the<br>presence of macules<br>(flat) and papules<br>(elevated). Also known<br>as morbillform rash, it is | symptoms (eg,<br>pruritus, burning,<br>tightness)<br>Erythema<br>covering <10%<br>BSA with or | (eg, pruritus,<br>burning, tightness);<br>limiting<br>instrumental ADL;<br>Erythema 30%<br>BSA with or | without<br>associated<br>symptoms;<br>limiting<br>self-care ADL | | |
| one of the most common cutaneous adverse events, frequently affecting the upper trunk, spreading centripetally, and associated with pruritus. | without<br>symptoms (eg,<br>pruritus, burning,<br>tightness) | without symptoms<br>(eg, pruritus,<br>burning, tightness);<br>limiting<br>instrumental ADL | Erythema<br>covering<br>> 30% BSA<br>with or<br>without<br>associated<br>symptoms;<br>limiting<br>self-careADL | | |

ADL = active daily living


# APPENDIX 7 PROTOCOL SUMMARY OF CHANGES

The protocol summary of changes was moved to the end of the protocol for easier readability.

Significant changes are described in the table below. Changed text is displayed for the first major occurrence only. Deleted text is presented in strikethrough format, and added text is presented in bold format.

| Section | <b>Description of Changes</b> | Rationale |
|---|---|---|
| Global | Replace: | Administrative |
| | Protocol Date and Version: 21 March 2018; V3.0 | |
| | With: | |
| Global | Change: | Administrative |
| | Changed Version number from V3.0 (Amendment 2) to V4.0 (Amendment 3) and Version date from 21 March 2018 to 27 July 2018. | |
| Global | Made administrative and editorial (formatting, typographical, and grammatical) updates. | Administrative |
| Global | Replaced subjects with <b>patients</b> . | Corrected wording used to refer to those participating in study with SLE. |
| Global | All references directly or contextually to MAD/POC "phase" or "study" have been replaced with "MAD portion/part/part of the study)" or "POC portion/part/part of the study". | Clarifies that MAD and POC are 2 portions of this 1 study and not 2 separate studies. |
| Global | When referring to the DMC and Boston Pharmaceuticals conducting a data review to determine POC dose, all instances of the phrase "suggest which dose should" have been replaced with "determine which dose will". | Protocol clarification. |
| Title Page | Replace: | Administrative |
| Appendix 1 | Boston Pharmaceuticals, Inc.<br>55 Cambridge Parkway, Suite 401<br>Cambridge, MA 02142 | |


### Section Description of Changes

Rationale

United States of America (USA)

With:

Boston Pharmaceuticals, Inc. 55 Cambridge Parkway, Suite 40**0** Cambridge, MA 02142 United States of America (USA)

CLINICAL PROTOCOL APPROVAL FORM Add: Administrative

PPD, MD, PhD
Chief Medical Officer
Boston Pharmaceuticals

Name and Title

PPD , MD, FACR Vice President, Clinical Development Boston Pharmaceuticals

CONFIDENTIALITY AND INVESTIGATOR STATEMENT

Replace:

I have read the protocol (V3.0 [Amendment 2], dated 21 March 2018), including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described.

With:

I have read the protocol (Version 4.0, dated **27 July** 2018), including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described.

PROTOCOL SUMMARY.

Background and Rationale

Replace:

The no observed adverse effect levels (NOAELs) in Cynomolgus monkeys were determined to be 100 mg/kg IV and 50 mg/kg SC, the highest doses tested. No SC animals had injection reactions.

With:

The no observed adverse effect level (NOAEL) in Cynomolgus monkeys was determined to be 100 mg/kg (SC and IV), the highest dose tested. There were no injection site reactions in animals dosed subcutaneously.

Updated based on new data describing NOAEL based on 6-month study data.

Administrative


#### BOS161721

#### Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 27 July 2018; V4.0 **Description of Changes** Section Rationale **PROTOCOL** Delete: Removed since this date SUMMARY, Background and Overall, there were no clinically significant safety or tolerability findings has been Rationale from this study, following an interim cut and review of the data at Day superseded. 90 postdose. Section 1.2.2.3, Clinical Studies PROTOCOL Delete: Removed as SUMMARY, not a safety Objectives and endpoint. Concomitant medication usage Endpoints, MAD Phase 1b, Safety Endpoints PROTOCOL SUMMARY, Objectives and Endpoints, POC Phase 2, Safety **Endpoints** Section 2.1, Phase 1b Multiple Ascending Dose, Safety **Endpoints** Section 2.2, Phase 2 Proof of Concept,

# PROTOCOL SUMMARY,

Objectives and Endpoints, MAD Phase 1b, Efficacy Endpoints

Safety Endpoints

Section 2.1, Phase 1b Multiple Ascending Dose, Efficacy Endpoints

#### Replace:



Statistical clarification.


**Description of Changes** Section Rationale





**PROTOCOL** SUMMARY,

Objectives and Endpoints, POC Phase 2, Secondary **Efficacy Endpoints** 

Section 2.2, Phase 2 Proof of Concept, Secondary Efficacy Endpoints

The proportion of **patients** with:

- SRI-4 response at each visit
- SRI-5 and SRI-6 response at each visit (Section 6.3.4.2)
- a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and  $\leq$  Day 0 dose) between Day 120 and Day 210
- new BILAG A flare or > 1 BILAG B flares relative to baseline through Day 210
- PGA worsening
- a BICLA response
- a CLASI response
- medication failures
- Results and changes from baseline in:
  - **CLASI**
  - swollen and tender joints ACR-28

Statistical clarification.


Section **Description of Changes** Rationale SLEDAI-2K SLICC/ACR damage index Time to medication failure Duration of **longest** SRI-4 response Time to first SRI-4 response Time to BILAG A flare or > 1 BILAG B flare compared to baseline through Day 210 PROTOCOL Replace: To include **SUMMARY**, Study more data Two weeks after the last patient in Cohort 3 receives the second dose, the from the Design DMC and Boston Pharmaceuticals will conduct a data review to suggest 120 mg cohort in data review which dose should be carried forward into the POC Phase 2 study. Section 1.2.4, Risk-Benefit to determine POC dose. Assessment With: Thirty days after the last patient in Cohort 3 receives the third dose, the DMC and Boston Pharmaceuticals will conduct a data review to determine which dose will be carried forward into the POC part of the study. Protocol PROTOCOL Add: SUMMARY, Study clarification. Design After successfully completing a screening phase, **eligible** patients will be randomized to a specified dose of BOS161721 or placebo. Section 3.1, Study Design PROTOCOL Add: Protocol SUMMARY, clarification. Inclusion Criteria 4 At screening, patients must have at least 1 of the following: Section 4.4, Inclusion a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the Criteria central laboratory Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory c. C3 or C4 levels below normal as determined by the central lab PROTOCOL Add: Protocol SUMMARY. clarification. **Exclusion Criteria** 9 Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically Section 4.5, significant is defined as requiring systemic parenteral antibiotics or Exclusion Criteria hospitalization 11 Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV) unless patient received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness


| Section | Description of Changes | | Rationale |
|---|---|---|---|
| PROTOCOL<br>SUMMARY,<br>Exclusion Criteria<br>Section 4.5,<br>Exclusion Criteria | Replace: 15 CD4+ count < 500/μL at screening With: 15 CD4+ count < 350/μL at screening | The cut off for plute count/µL culating levels in current trial is a Erythematosus disease, are enia and dispenia with 00 cells/µL. case definitions and revised unological ated disease in 4+ count a classified as dency, thus the d for exclusion 4+ cells/ µL. | |
| PROTOCOL<br>SUMMARY,<br>Exclusion Criteria<br>Section 4.5,<br>Exclusion Criteria | Delete: 17 Hemoglobin < 8 g/dL or < 7 g/dL at screen related to SLE | Text removed<br>as lab values<br>would already<br>qualify as<br>anemic. | |
| PROTOCOL<br>SUMMARY,<br>Statistical<br>Considerations | dose based on Phase 1 data, and 2) a final analy Additionally, DMC safety analyses will be perf cohort and throughout Phase 2 to monitor patient Unless stated otherwise, statistical testing will of Phase 2 data and will be done using 2-sided over With: Two analyses are planned: 1) an interim analyses | Two analyses are planned: 1) an interim analysis to select the Phase 2 dose based on Phase 1 data, and 2) a final analysis at study completion. Additionally, DMC safety analyses will be performed after each Phase 1 cohort and throughout Phase 2 to monitor patient safety. Unless stated otherwise, statistical testing will only be performed on the Phase 2 data and will be done using 2-sided overall alpha of 0.10. With: | |
| | based on the MAD data, and 2) a final analysis Additionally, DMC safety analyses will be perf cohort and throughout the POC to monitor pati the DMC charter. Unless stated otherwise, statistical testing will composed poor and will be done using 2-sided overall. | formed for each MAD eent safety as described in only be performed on the | changes and<br>additions to<br>provide<br>further clarity<br>to Phase 1 and<br>2 being MAD<br>and POC. |
| Section 1.2.2,<br>BOS161721<br>Development | Add: Boston Pharmaceuticals is developing BOS161 SLE. BOS161721 is a humanized immunoglob extended half-life directed against human IL-2 | oulin G1 (IgG1) mAb with | Protocol clarification. |


#### Section

#### **Description of Changes**

#### Rationale

#### Section 1.2.2,2 Preclinical Studies

Replace:

The NOAELs were determined to be 100 mg/kg IV and 50 mg/kg SC, the highest doses tested.

With:

Updated based on new data describing NOAEL based on 6-month study data.

The NOAEL was determined to be 100 mg/kg (SC and IV), the highest dose tested.

#### Section 1.2.2,2 Preclinical Studies

Add:

An additional GLP, repeat-dose toxicity study was conducted in Cynomolgus monkeys (4 males and 4 females per dose group) following every 2 weeks (Q2W) administration by SC (10, 30, and 100 mg/kg) injection for a total of 14 doses.

There were no BOS161721-related effects on

Data from a 6 month GLP Toxicology study conducted in Cynomolgus monkeys was not available at the time the original protocol was written.

There were no BOS161721-related effects on survival, clinical signs, male body weights, ophthalmologic parameters, electrocardiogram (ECG) findings, clinical pathology, macroscopic observations, organ weights, or microscopic



Section 1.2.3, Study Dose Selection Add:

Protocol clarification.

Doses have been selected for the multiple ascending dose (MAD) Phase 1b portion based on a 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01); the SDMT reviewed the blinded safety data from subjects for each dose cohort (8 cohorts, evaluating 1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg), along with the accumulated safety and available PK/PD data from all subjects in the previous dose cohorts, to make a decision on whether to proceed to the next higher dose level, repeat a dose level, or stop dose escalation.


#### Section **Description of Changes** Rationale Section 1.2.5. Protocol Delete: Potential Risks clarification. ADAs could result in immune complex disease (with manifestations such as arthralgias, serum-sickness, and vasculitis), autoimmunity, or altered BOS161721 levels or activity. Section 1.2.5.2, Replace: Data was not Injection Site available at Reactions In a repeat-dose GLP toxicology study in Cynomolgus monkeys, the time the BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) for original 3 months (a total of 7 doses); no SC animals had injection reactions. protocol was written. With: In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC for 3 months (a total of 7 doses). There were no injection site reactions in animals

dosed subcutaneously. Further, there were no reports of injection site reactions in the 26-week GLP toxicology study in Cynomolgus

# Section 1.2.5.4, Infections

#### Replace:

monkeys.

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells,<sup>37</sup> patients with a CD4+ count < 500 cell/mm<sup>3</sup> were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from the proposed MAD/POC studies.

#### With:

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells,<sup>37</sup> patients with a CD4+ count < 500 cell/mm<sup>3</sup> were excluded from the Phase 1 SAD study (BOS161721-01), and **CD4** + < **350** cells/mm<sup>3</sup> will be excluded from the MAD/POC parts of the study.

DMC recommendation: The cut off for CD4+ T cells of 500 absolute count/µL was based on normal circulating levels in healthy individuals. The current trial is enrolling Systemic Lupus Erythematosus patients that, due to the disease, are known to have lymphopenia and specifically CD4+ lymphopenia with values typically below 500 cells/µL. According to the "WHO case definitions of HIV for surveillance and revised clinical staging and immunological classification of HIV-related disease in adults and children". CD4+ count  $< 350 \text{ cell/}\mu\text{L in}$ adults is classified as significant immunodeficiency, thus the proposed cutoff threshold for exclusion criteria will be  $< 350 \text{ CD4+ cells/}\mu\text{L}$ .


#### Section Description of Changes

#### Section 1.2.5.6, Hepatic Function

Abnormality

#### Replace:

However, as a precaution, patients with a history of abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST  $> 2 \times$  upper limit of normal [ULN]; total bilirubin  $> 1.5 \times$  [ULN] and judged by the investigator to be clinically significant) were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from the MAD study.

#### With:

However, as a precaution, patients with a history of abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST  $> 2 \times$  upper limit of normal [ULN]; total bilirubin  $> 1.5 \times$  [ULN] and judged by the investigator to be clinically significant) were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from **this trial**.

# Section 3.1, Study Design

#### Replace:

The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease being studied.

#### With:

The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease **activity**.

#### Section 3.1.1, Multiple Ascending Dose Phase 1b Study

#### Add:

All doses selected for the MAD **part of the** study are projected not to exceed the mean exposure of that achieved in the SAD study.

# Section 3.1.1.3, DMC Recommendations

#### Replace:

The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available at the time the last patient in Cohort 3 completes the Day 44 visit (2 weeks after dose 2).

#### With:

The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available 30 days after the last patient from Cohort 3 receives the third dose.

#### Rationale

Protocol clarification -MAD and POC have the same entrance criteria.

Protocol clarification.

Protocol clarification.

To include more data from the 120 mg cohort in data review to determine the POC dose.


| Section | Description of Changes | Rationale |
|---|---|---|
| Section 3.1.2.1,<br>BOS161721 Dose | Delete: The optimal dose evaluation is chosen based on MAD Phase 1b safety, | Protocol clarification. |
| | tolerability, immunogenicity, and PK and PD data. | |
| Section 3.2,<br>Randomization and | Replace: | Protocol clarification. |
| blinding, Table footnote | *Additional patients may be enrolled to confirm sufficient numbers of patients are in the full analysis set (FAS). | |
| | With: | |
| | *Additional patients may be enrolled to <b>ensure</b> sufficient numbers of patients are in the full analysis set (FAS). | |
| Section 3.2,<br>Randomization and | Add: | Protocol clarification. |
| blinding | Similarly, patients in the Phase 1b MAD will be assigned to the cohort which is active. | ciaiiiication. |
| Section 3.3, Study<br>Schematic | Replace: | Protocol clarification. |

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2 Studies



With:

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2




#### Section

#### **Description of Changes**

#### Section 3.4, Schedule of Assessments, Table 1, Safety Follow-Up column

Add:

| | Safety Follow-Up | | |
|---|---|---|---|
| Days | 210 (± 3) | 240 (± 3) | 270 (± 3) |
| Visit Number | 11 | 12 | 13 |
| Urine pregnancy<br>test (women) <sup>n</sup> | | | X |

Protocol clarification. Urine pregnancy test added at day 270 to ensure patient is not pregnant at end of 90 day follow-up due to 41 day half-life of study drug. Adding PK windows for added flexibility.

Rationale

Section 3.4, Schedule of Assessments, Table 1, PK Labs Windows

Add:

| | Screen <sup>a</sup> | Enroll | | | | Tr | eatment | Period 1 | Follow-I | Jp . | | | 500000 B | Safet | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28<br>to -1 | 0 | 7<br>(±1) | 15<br>(± 3) | 30<br>(± 3) | 44<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit number | 1 | 2 | ** | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | ** | - | 11 | 12 | 13 |
| PK Labs | | | | | | - | | | | | | | | | | |
| Predose | | X | | | X | | X | X | X | X | X | | | | | |
| Predose PK<br>Window | | 60m | | | ± 3d | | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | | | | | |
| Postdose | | XP | X | X | ΧP | | | | | | Χ» | X | X | X | X | X |
| Postdose PK<br>Window | | 4h ±<br>30m<br>8h ±<br>45m<br>24h ±<br>60m | ± 1d | ± 3d | 4h ±<br>30m<br>8h ±<br>45m<br>24h ±<br>60m | | | | | | 4h ±<br>30m<br>8h ±<br>45m<br>24h ±<br>60m | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d |

Protocol clarification.

Section 3.4, Schedule of Assessments, Table 1 footnotes

Add:

Section 3.4, Schedule of Assessments, Table 2 footnotes

Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed (analyzed) if the patient had a positive ADA on Day 90.

Protocol

clarification.

Section 3.4, Schedule of Assessments.

Table 1 footnotes

nAb is assessed if patient is positive for ADA.

Section 3.4, Schedule of Assessments,

Table 2 footnotes

nAb is collected for all patients, though will only be analyzed by central lab if patient is positive for ADA at Day 90.

Section 3.4, Schedule of Assessments, Table 1 footnotes

Add:

With:

Replace:

collected during safety follow-up visits. Only CC

Protocol clarification.

 BOS161721 Boston Pharmaceuticals, Inc.


#### Section

#### **Description of Changes**

#### Section 3.4, Schedule of Assessments, Table 2 Safety Follow-Up column

Add:

| | Safety Follow-Up | | |
|---|---|---|---|
| Days | 210 (± 3) | 240 (± 3) | 270 (± 3) |
| Visit Number | 10 | 11 | 12 |
| Urine pregnancy test (women) <sup>m</sup> | | | X |

Rationale

Protocol clarification urine pregnancy test added at day 270 to ensure patient is not pregnant at end of 90 day follow-up due to 41 day half-life of study drug. Adding PK windows for added flexibility.

Section 3.4, Schedule of Assessments, Table 2, PK Labs Window Add:

| | Screen <sup>a</sup> | reen* Enroll Treatment Period Follow-up | | | | | | Safety Follow-Up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28 to -1 | 0 | 15<br>(± 3) | 30<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(±3) | 270<br>(±3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | - | 10 | 11 | 12 |
| PK Labs* | | | | - | | | - | | | | | | - | |
| Predose | | X | | X | X | X | X | X | X | | | | | |
| Predose PK Window | | 60m | | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | | | | | |
| Postdose | | 30.00 | X | | | - 6-1 | - | | | X | X | X | X | X |
| Predose PK Window | | | ± 3d | | | | | | | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d |

Section 3.4, Schedule of Assessments, Table 2 footnotes

Add:

Only CCI collect

collected during safety follow-up visits.

Protocol clarification.

Section 3.5, End of Study

Add:

#### 3.5 End of Study

End of Study (Individual Patient): A patient is considered at the end of study if he/she has withdrawn, prematurely discontinued, or completed all of the study procedures including the last visit.

End of Study (End of trial): The end of the study is defined as the date of the last visit of the last patient in the study globally, or the date of which the last patient withdraws or discontinues if all prior enrolled patients have already completed/withdrawn.

Added end of study definitions in alignment with recent agency protocol authoring guidance.

Section 4.6.2, Other Prohibited and/or Restricted Treatments Replace:

- Patients who have received treatment with anti-CD20 monoclonal antibodies within 6 months of screening; recovery of B cells (CD19+) must be documented (record absolute number of CD19+ B cells)
- Patients who have received treatment with cyclophosphamide within the 1 year prior to screening
- 4 Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria (oral or topical) within 3 months of screening
- 5 Patients who are currently receiving or are scheduled to receive

Protocol clarification to align with appendices, align with other windows in protocol, and further clarification in #4 for sites to differentiate between oral and topical washout.


BOS161721 Boston Pharmaceuticals, Inc.


#### Section Description of Changes Rationale

plasmapheresis or lymphapheresis therapy, or have received such therapy within 8 weeks prior to screening

#### With:

- Patients who have received treatment with anti-CD20 monoclonal antibodies within **24 weeks** of screening; recovery of B cells (CD19+) must be documented (record absolute number of CD19+ B cells)
- Patients who have received treatment with cyclophosphamide within the **24 weeks** prior to screening
- 4 Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria within 4 weeks for oral use or 8 weeks for topical use of screening
- 5 Patients who are currently receiving or are scheduled to receive plasmapheresis or lymphapheresis therapy, or have received such therapy within 24 weeks prior to screening

#### Section 5.1, Screening

Add:

Protocol clarification.

• Chest x-ray (a prior x-ray can be used if taken within 12 weeks of screening date)

#### Section 5.2, Enrollment/

Randomization and Day 0 Treatment

Replace:

The study site will obtain a randomization number when registering the patient in IWRS.

Added text to ensure eligibility prior to randomization

With:

Prior to randomization, the study site should confirm that the patient still meets inclusion/exclusion criteria (especially SLE disease activity and treatment). The site will obtain a randomization number when registering the patient in IWRS.

## Section 5.3,

Treatment Period/Follow-Up Visits Replace:

Protocol clarification.

• CRP and nAb will be assessed if patient is positive for ADA

#### With:

- nAb will be analyzed by central lab if patient is positive for ADA
- CRP


BOS161721


| Section | Description of Changes | Rationale |
|---|---|---|
| Section 5.4, Safety<br>Follow-Up Visits | Add: | Urine pregnancy test |
| | • Urine pregnancy test | added at day 270 to ensure patient is not pregnant at end of 90 day follow up due to 41 day half-life of study drug. |
| Section 6.2.1, | Delete: | Central data is not being |
| Laboratory<br>Assessments | A central laboratory will be used (with the exception of urine pregnancy tests-and stool analysis) to ensure accuracy and consistency in test results. The central laboratory will transmit all results for protocol tests, scheduled and unscheduled, to the clinical data base. | transmitted into the clinical database. |
| Section 6.2.1, | Add: | Protocol |
| Laboratory Assessments, Table 3, | Other Safety Tests | clarification to align with |
| Other Safety Tests column | Spot urine for protein/creatinine ratio FSH <sup>b</sup> | Schedule of Assessments. |
| | Urine pregnancy test <sup>c</sup> QuantiFERON®-TB Gold In-Tube test (QFT-G) <sup>d</sup> Serology <sup>d</sup> (Hepatitis B and C; HIV-1/2 combination) Stool sample <sup>c</sup> Serum pregnancy test | |
| Section 6.2.1, | Add: | Protocol |
| Laboratory Assessments, Table 3, Additional Tests | Additional Tests <sup>f</sup> | clarification to<br>align with<br>Schedule of |
| column | (potential Hy's Law) AST, ALT (repeat) Total bilirubin (repeat) Albumin (repeat) Alkaline phosphatase (repeat) Direct bilirubin | Assessments. |
| | Indirect bilirubin GGT Prothrombin time/international normalized ratio (repeat) | |
| S-4 (2.1.1 | Creatine kinase (repeat) | II.i |
| Section 6.2.1.1, Pregnancy Testing | Add: Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, at the last follow up visit day (Day 270) and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. | Urine pregnancy test added at day 270 to ensure patient is not pregnant at end of 90 day follow up due to 41 day half-life of |


Clinical Study Protocol: BOS161721-02
Section Description of Changes

| Section | Description of Changes | Rationale |
|---|---|---|
| Section 6.2.2.2,<br>Recording of Adverse<br>Events | Delete: The details of the AE, date of AE onset (and time, if known), date of AE outcome (and time, if known), and action taken for the AE will be documented together with the principal investigator's assessment of the seriousness of the AE and causal relationship to the study drug and/or the study procedure. | Exact time of adverse event is not needed for this study. If serious adverse event, time of onset will be provided in narrative. |
| Section 6.2.2.6.2,<br>Injection Site<br>Reactions | Add: These will include Grades 2 to 5 injection site erythema, pain, and induration (see APPENDIX 6), which are also captured as Adverse Events of Special Interest (See Section 6.2.2.6). | Protocol clarification. |
| Section 6.2.3, Vital Signs | Add: Vital signs will be assessed on Day 0 at predose and at <b>Day 0</b> , 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). | Protocol clarification. |
| Section 6.2.8,<br>Immunogenicity | Replace: Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90. After the first dose, if a patient tests positive in the validated confirmatory ADA assay, the sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay. With: Subsequent ADA samples will be collected from all patients but only analyzed by a central lab if the patient had a positive ADA on Day 90. After the first dose, if a patient tests positive in the validated confirmatory ADA assay, a sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay by a central lab. | Protocol clarification. |
| Section 6.3.3, PGA of Disease Activity | Add: PGA worsening is defined as an increase of > 30 mm from baseline. | Added definition of worsening PGA. |
| Section 6.3.4.1, SRI-4<br>Response | Replace: no deterioration from baseline in the PGA by $\geq 0.3$ points With: no deterioration from baseline in the PGA by $\geq$ 30 mm | Unit was incorrectly presented in previous protocol version. |


| Section | Description of Changes | Rationale |
|---|---|---|
| Section 6.3.4.2, SRI-5 and SRI-6 Response | Replace: However, the SRI-5 and SRI-6 are computed with a minimal three-point or five point improvement in SLEDAL 2V being required representatively. | Units incorrectly presented in previous |
| | or five-point improvement in SLEDAI-2K being required, respectively. With: | protocol version. |
| | with. | version. |
| | However, the SRI-5 and SRI-6 are computed with a minimal <b>five</b> -point or <b>six</b> -point improvement in SLEDAI-2K being required, respectively. | |
| Section 6.4.2, PROs | Add: | Protocol clarification. |
| | CCI | ciarrication. |
| Section 8, Statistics | Add: | Protocol clarification. |
| | • The final analysis will be performed when all patients have completed the <b>POC</b> safety follow-up or withdrawn from the study. | Charmeanon. |
| Section 8, Statistics | Replace: | If an interpolated |
| | Select parameters will be summarized using patients from both study phases. | dose is selected for POC, dose |
| | With: | levels may not be combined. |
| | Select parameters <b>may</b> be summarized using patients from both study <b>parts</b> . | |
| Section 8.2.3, Primary Efficacy Endpoint(s) | Delete: | Statistical inference will |
| Efficacy Enapoliti(s) | If the proportion of SRI-4 responders for the selected POC dose in BOS161721 arm is higher than that of the placebo arm, then BOS161721 will be considered superior to placebo if the 2-sided p-value is less than or equal to-0.10. | be based on a<br>2-tailed test<br>with an overall<br>0.10 level of<br>significance. |
| Appendix 1 | Replace: | Administrative |
| | PPD | |
| | PPD | |
| | With: | |
| | PPD | |


| Section | Description of Changes | Rationale |
|---|---|---|
| | PPD | |
| | PPD | |
| | PPD | |
| Appendix 4 | Add: | Protocol clarification. |
| | Cyclosporine (except for CSA eye drops) 4 weeks for oral and 8 weeks topical | for |




## A RANDOMIZED DOUBLE-BLIND PHASE 1b/2 COMBINED STAGGERED MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF LIMITED STANDARD OF CARE

**SPONSOR** Boston Pharmaceuticals, Inc.

55 Cambridge Parkway, Suite 401

Cambridge, MA 02142

United States of America (USA)

INVESTIGATIONAL COMPOUND: BOS161721

PROTOCOL NUMBER: BOS161721-02

PHASE Phase 1b/2

INVESTIGATIONAL NEW DRUG (IND) 131796

**NUMBER:** 


**VERSION NUMBER:** V3.0 (Amendment 2)

**VERSION DATE:** 21 March 2018

BOS161721

Clinical Study Protocol: BOS161721-02


## CLINICAL PROTOCOL APPROVAL FORM

Protocol Title: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

Study No: BOS161721-02

Original Protocol Date: 06 October 2017 Protocol Version No: v2.0 (Amendment 1) Protocol Version Date: 14 November 2017 Protocol Version No: v3.0 (Amendment 2) Protocol Version Date: 21 March 2018

This study protocol was subject to critical review and has been approved by sponsor. The information contained in this protocol is consistent with:

- The current risk-benefit evaluation of the investigational product.
- The moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (APPENDIX 2), and principles of Good Clinical Practices (GCP) as described in 21 Code of Federal Regulations (CFR) parts 50, 54, 56 and 312 and according to applicable local requirements.

The investigator will be supplied with details of any significant or new findings, including adverse events, relating to treatment with the investigational product.

I agree with these statements and indicate my approval by signature for this protocol:

| Name and Title | Signature and Date |
|---|---|
| PPD , MD Vice President, Clinical Development Boston Pharmaceuticals | PPD |
| PPD Clinical Operations Lead Boston Pharmaceuticals | PPD |
| PPD , MD, PhD Vice President, Clinical Development and Safety Officer Boston Pharmaceuticals | PPD |


BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02 Protocol Date and Version: 21 March 2018; V3.0

#### BOS161721-02

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

## CONFIDENTIALITY AND INVESTIGATOR STATEMENT

The information contained in this protocol and all other information relevant to BOS161721 are the confidential and proprietary information of Boston Pharmaceuticals, Inc., and except as may be required by federal, state, or local laws or regulation, may not be disclosed to others without prior written permission of Boston Pharmaceuticals, Inc.

I have read the protocol (V3.0 [Amendment 2], dated 21 March 2018), including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described. I will conduct this study as outlined herein, in accordance with the regulations stated in the Federal Code of Regulations for Good Clinical Practices and International Council for Harmonisation (ICH) guidelines, and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and any amendments, and access to all information provided by Boston Pharmaceuticals, Inc., or specified designees. I will discuss the material with them to ensure that they are fully informed about BOS161721 and the study.

| Principal 1 | Investigator Name (printed) | Signature |
|-------------|----------------------------------------|-----------|
| ————Date | —— ——————————————————————————————————— | |


# PROTOCOL SUMMARY

| Title: | A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care |
|---|---|
| Indication | Adults with moderately to severely active SLE |
| Background and Rationale | SLE is a chronic systemic autoimmune disease with considerable heterogeneity in clinical manifestations and disease course. There is evidence that B- and T-cells are critical to the development of the disease, and that T-cell-derived cytokines such as interleukin-21 (IL-21) are involved in the SLE-associated inflammatory pathological response. |
| | BOS161721 is a humanized immunoglobulin G1 (IgG1) triple mutation monoclonal antibody (mAb) intended to have an extended terminal elimination half-life (t <sub>1/2</sub> ) that selectively binds to and neutralizes IL-21, which acts on multiple cell types that drive inflammation and autoimmunity. In vivo, BOS161721 inhibits T-cell dependent antigen responses of B-cells and is being developed as a potential treatment for adults with moderately to severely active SLE. |
| | Nonclinical studies have evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), pharmacokinetics (PK), and immunogenicity of BOS161721 administered intravenously (IV) and subcutaneously (SC). The no observed adverse effect levels (NOAELs) in Cynomolgus monkeys were determined to be 100 mg/kg IV and 50 mg/kg SC, the highest doses tested. No SC animals had injection reactions. |
| | In a Phase 1 single ascending dose (SAD) study, BOS161721 was administered IV and SC to healthy male and female adult subjects. This double-blind, placebo-controlled study evaluated 8 ascending dose levels (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) for safety, tolerability, PK, PD and immunogenicity. Overall, there were no clinically significant safety or tolerability findings from this study, following an interim cut and review of the data at Day 90 postdose. |
| | Results from the Phase 1 SAD study informed the dose regimens used for the multiple ascending doses (MAD) Phase 1b study in this trial. The MAD study will involve 3 cohorts. The Phase 2 portion will be a proof of concept (POC) study, where dose selection will be based on the data monitoring committee (DMC) and sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD study of 30 patients treated with BOS161721/placebo. The purpose of the study is to establish safe and effective dosages for adult patients with moderately to severely active SLE. |


## **Objectives and Endpoints:**

## **MAD Phase 1b Study**

#### **OBJECTIVES ENDPOINTS** Primary To assess safety, tolerability, and Safety Endpoints immunogenicity of repeat doses of Incidence and severity of adverse events BOS161721 (20, 60, and 120 mg) (AEs) and serious adverse events (SAEs), administered SC in adult patients related AEs, AEs leading to study drug with moderately to severely active discontinuation, AEs by severity and SLE on limited background relatedness standard of care treatment, in order Injection site reactions to estimate the optimal dose. Columbia Suicide severity Rating Scale 12-lead electrocardiograms (ECGs) parameter results at each visit and change from baseline Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline Clinical laboratory results and change from baseline Physical examinations changes from baseline Anti-drug antibodies (ADAs) Study drug exposure/compliance Concomitant medication usage Secondary To characterize the PK of Pharmacokinetic Endpoints BOS161721 and select the optimal BOS161721 concentration by visit and time dose of BOS161721 based on safety, PK, and PD effects in Maximum observed concentration (C<sub>max</sub>), patients with mild to moderate first time to maximum concentration (T<sub>max</sub>), SLE. area under the concentration-time curve (AUC), $t_{1/2}$ , systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>) Pharmacodynamic Endpoints Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit Results and changes (or shifts) from baseline in abrogation of IL-21 gene

signature at each indicated visit

Exploratory



# **POC Phase 2 Study**

| OBJECTIVES | ENDPOINTS |
|------------|-----------|
| Primary | |

BOS161721 Boston Pharmaceuticals, Inc.


> To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on the SLE Responder Index 4 (SRI-4)

## Primary Efficacy Endpoint

The proportion of subjects with a SRI-4 response at Day 210 (see Section 6.3.4.1)

#### **Secondary**

 To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment

#### Secondary Efficacy Endpoints

- The proportion of subjects with:
  - SRI-4 response at each visit
  - SRI-5 and SRI-6 response (Section 6.3.4.2)
  - a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210
  - new BILAG A flare or > 1 BILAG B flares relative to baseline through Day 210
  - PGA worsening
  - a BICLA response
  - a CLASI response
  - medication failures
- Results and changes from baseline in:
  - CLASI
  - swollen and tender joints ACR-28
  - SLEDAI-2K
  - SLICC/ACR damage index
  - Time to medication failure
- Duration of SRI-4 response
- Time to first SRI-4 response
- Time to BILAG A flare or > 1 BILAG B flare compared to baseline through Day 210

#### Safety

BOS161721


> To assess safety and tolerability of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment

#### Safety Endpoints

- Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness
- Injection site reactions
- C-SSRS
- 12-lead ECGs parameter results at each visit and change from baseline
- Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline
- Clinical laboratory results and change from baseline
- Physical examinations changes from baseline
- ADAs
- Study drug exposure/compliance

Concomitant medication usage



#### **Study Design:**

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of multiple SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly. The trial will consist of 2 double-blinded studies: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90,

120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

The MAD Phase 1b study phase will consist of 3 cohorts, with Cohort 1 containing 6 patients, where 5 of these patients will receive BOS161721 (active), and 1 will receive placebo. Cohorts 2 and 3 will each contain 12 patients, including 9 active and 3 placebo patients. Dose selection for each cohort is based on 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. Each of the 3 doses (20, 60, and 120 mg) selected for the MAD study are projected not to exceed the mean exposure of that achieved in the SAD study following the single 240 mg SC dose. Each patient may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

The MAD study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after a DMC evaluates the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after DMC evaluation of the safety and tolerability data from Cohort 2 and Cohort 1. Two weeks after the last patient in Cohort 3 receives the second dose, the DMC and Boston Pharmaceuticals will conduct a data review to suggest which dose should be carried forward into the POC Phase 2 study. This dose will not exceed doses tested during the MAD study.

For the POC study, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio. As in the MAD study, each patient in the POC study may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 60. Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits. Tapering may occur after randomization except within 60 days of the primary (Day 210) and secondary (Day 120) endpoint assessments. Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant.

DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.

# Main Criteria for Inclusion

#### **Inclusion Criteria:**

#### and Exclusion

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion OR Lupus nephritis as the sole clinical criterion in the presence of antinuclear antibodies [ANA] or anti- double-stranded deoxyribonucleic acid [dsDNA] antibodies), either sequentially or simultaneously
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
  - c. C3 or C4 below normal as determined by the central lab
- 5. At screening, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia
    - ii. Points from lupus headache and organic brain syndrome will also

#### be excluded

- 7. Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 4.4

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization)
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of

sperm turnover) for a total of 44 weeks after treatment completion

11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

#### **Exclusion Criteria**

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed

8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study

- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count < 500/μL at screening
- 16. Platelets < 50,000/mm<sup>3</sup> (50  $\times$  10<sup>9</sup>/L) or < 35,000/ mm<sup>3</sup> (35  $\times$  10<sup>9</sup>/L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if due to anemia related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation
- 20. Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) > 2 × the upper limit of normal (ULN) at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK) > 3.0 × ULN at screening unless related to lupus myositis
- 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic mAb (eg, IgG protein) or molecules made of components of mAbs
- 25. History substance and/or alcohol abuse, or dependence within the past 1 year, at the investigator's judgment

26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision

- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 on the C-SSRS
- 31. Current or pending incarceration
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness

# Statistical Considerations

Below is a summary of the statistical methods. Further details can be found in Section 8.

Two analyses are planned: 1) an interim analysis to select the Phase 2 dose based on Phase 1 data, and 2) a final analysis at study completion. Additionally, DMC safety analyses will be performed after each Phase 1 cohort and throughout Phase 2 to monitor patient safety.

Unless stated otherwise, statistical testing will only be performed on the Phase 2 data and will be done using 2-sided overall alpha of 0.10. Data will be summarized descriptively by treatment and overall for each study phase. For the MAD phase, BOS161721 will be summarized overall and by each dose level and placebo patients from each cohort will be combined.

The descriptive summaries for the categorical data will include number and percentage. The descriptive summaries for the continuous data will include number, mean, median, standard deviations (SD), 25th and 75th percentiles, minimum, median, and maximum. Counts, medians, 25th and 75th percentiles, and standard error will be presented for time-to-event data.

All safety analyses will be performed using the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. All efficacy analyses will be performed using the full analysis set (FAS), defined

as all patients who receive at least 1 dose of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. Select efficacy analyses may also be performed on the per protocol (PP) set.

Binary efficacy endpoints, including the primary efficacy endpoint, will be assessed via Pearson's chi-squared analysis.

Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) when applicable, adjusting for the baseline value. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test.

Adverse event data will be coded to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be summarized, based on coded terms, using frequency and percentage of patients. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters, will be summarized at each individual visit.

# TABLE OF CONTENTS

| TITLE PAGE | 1 |
|----------------------------------------------------|----|
| CLINICAL PROTOCOL APPROVAL FORM | 2 |
| CONFIDENTIALITY AND INVESTIGATOR STATEMENT | 3 |
| PROTOCOL SUMMARY | 4 |
| TABLE OF CONTENTS | 16 |
| LIST OF IN-TEXT TABLES | 19 |
| LIST OF IN-TEXT FIGURES | 19 |
| LIST OF ABBREVIATIONS | 20 |
| 1. INTRODUCTION AND RATIONALE | 24 |
| 1.1 Indication | 24 |
| 1.2 Background and Rationale | 24 |
| 1.2.1 Overview of the Disease State | 24 |
| 1.2.2 BOS161721 Development | |
| 1.2.2.1 Interleukin-21 | 25 |
| 1.2.2.2 Preclinical Studies | 26 |
| 1.2.2.3 Clinical Studies | 27 |
| 1.2.3 Study Dose Selection | 28 |
| 1.2.4 Risk-Benefit Assessment | 29 |
| 1.2.5 Potential Risks | 29 |
| 1.2.5.1 Anaphylaxis and Serious Allergic Reactions | 30 |
| 1.2.5.2 Injection Site Reactions | 30 |
| 1.2.5.3 Immune Complex Disease | 31 |
| 1.2.5.4 Infections | 31 |
| 1.2.5.5 Malignancy | 32 |
| 1.2.5.6 Hepatic Function Abnormality | 32 |
| 1.2.5.7 Failure of Vaccination | 33 |
| 1.2.5.8 Potential for Drug-Drug Interactions | 33 |
| 1.2.5.9 Potential Risk to Fetal Development | 33 |
| 2 STUDY OBJECTIVES AND ENDPOINTS | 33 |
| 2.1 Phase 1b Multiple Ascending Dose | 34 |
| 2.2 Phase 2 Proof of Concept | 35 |
| 3 STUDY PLAN | 37 |
| 3.1 Study Design | 37 |
| 3.1.1 Multiple Ascending Dose Phase 1b Study | 37 |
| 3.1.1.1 Dose Escalation for the MAD Study | 38 |
| 3.1.1.2 Dose Limiting Toxicity (DLT) | 38 |
| 3.1.1.3 DMC Recommendations | 39 |

| Clinical Study Protocol: | BOS161721-02 |
|--------------------------|--------------|
|--------------------------|--------------|

|-------------------|----------|----------|-------|------|
|-------------------|----------|----------|-------|------|

| 3.1.2 | POC Phase 2 Study | 39 |
|---------|-------------------------------------------------------------|----|
| 3.1.2.1 | BOS161721 Dose | 39 |
| 3.1.2.2 | POC Study Design | 39 |
| 3.2 | Randomization and Blinding | 40 |
| 3.3 | Study Schematic | 41 |
| 3.4 | Schedule of Assessments | 42 |
| 4 PC | PULATION | 50 |
| 4.1 | Participant Recruitment | 50 |
| 4.2 | Number of Patients | 50 |
| 4.3 | Patient Screening | 50 |
| 4.4 | Inclusion Criteria | 50 |
| 4.5 | Exclusion Criteria | 52 |
| 4.6 | Concomitant Medications | 54 |
| 4.6.1 | Oral Corticosteroid Dose | 55 |
| 4.6.2 | Other Prohibited and/or Restricted Treatments | 56 |
| 4.7 | Women of Childbearing Potential | 56 |
| 4.7.1 | Determination of Menopause | 56 |
| 4.7.2 | Contraception | 57 |
| 4.8 | Deviation from Inclusion/Exclusion Criteria | 57 |
| 4.8.1 | Patient Withdrawal and Replacement | 58 |
| 5 ST | UDY PROCEDURES | 58 |
| 5.1 | Screening. | 58 |
| 5.1.1 | Retesting During Screening Period | 59 |
| 5.2 | Enrollment/Randomization and Day 0 Treatment | 59 |
| 5.3 | Treatment Period/Follow-Up Visits | 60 |
| 5.4 | Safety Follow-Up Visits | 61 |
| 5.5 | Premature Discontinuation. | 62 |
| 6 AS | SSESSMENTS | |
| 6.1 | Medical History, Demographic and Other Baseline Information | 62 |
| 6.2 | Safety Assessments | 63 |
| 6.2.1 | Laboratory Assessments | 63 |
| 6.2.1.1 | Pregnancy testing | 65 |
| 6.2.1.2 | Tuberculosis Screening | 65 |
| 6.2.2 | Adverse Events | 66 |
| 6.2.2.1 | Definitions | 66 |
| 6.2.2.2 | Recording of Adverse Events | 66 |
| 6.2.2.3 | Severity of Adverse Events | 66 |
| 6.2.2.4 | Causality of Adverse Events | 67 |
| 6.2.2.5 | Seriousness of Adverse Events | 67 |
| 6.2.2.6 | Adverse Events of Special Interest | 68 |
| 6.2.2.7 | Reporting of Adverse Events | 71 |

| Clinical Study Protocol: | BOS161721-02 |
|--------------------------|--------------|
|--------------------------|--------------|

|-------------------|----------|----------|-------|------|
|-------------------|----------|----------|-------|------|

| 6.2.2.8 | Follow Up of Adverse Events | 73 |
|---------|--------------------------------------------------------------|----|
| 6.2.3 | Vital Signs | |
| 6.2.4 | 12-Lead Electrocardiograms | 73 |
| 6.2.5 | Physical Examinations | 73 |
| 6.2.6 | C-SSRS | 74 |
| 6.2.7 | Injection Site Reactions | 74 |
| 6.2.8 | Immunogenicity | 74 |
| 6.3 | Efficacy Assessments | 75 |
| 6.3.1 | SLEDAI-2K | 75 |
| 6.3.2 | BILAG 2004 | 75 |
| 6.3.3 | PGA of Disease Activity | 75 |
| 6.3.4 | Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response | 76 |
| 6.3.4.1 | SRI-4 Response | 76 |
| 6.3.4.2 | SRI-5 and SRI-6 Response | 76 |
| 6.3.4.3 | BICLA Response | 76 |
| 6.3.5 | CLASI Response | 76 |
| 6.3.6 | ACR-28 Joint Count | 76 |
| 6.4 | Other Variables | 77 |
| 6.4.1 | SLICC/ACR Damage Index | 77 |
| 6.4.2 | PROs | |
| 6.5 | Pharmacokinetic Assessments | 77 |
| 6.6 | Pharmacodynamic Assessments | 77 |
| 6.7 | Pharmacokinetic/Pharmacodynamic Relationship | 78 |
| 6.8 | Protocol Deviations. | |
| 7 ST | ΓUDY DRUG MANAGEMENT | 78 |
| 7.1 | Description | 78 |
| 7.1.1 | Formulation | 78 |
| 7.1.2 | Storage | 78 |
| 7.2 | Packaging and Shipment | 78 |
| 7.3 | Dose and Administration | 78 |
| 7.4 | Accountability | 79 |
| 7.5 | Prohibited Concomitant Therapy | 79 |
| 7.6 | Compliance | 79 |
| 8 S7 | TATISTICS | 79 |
| 8.1 | Sample Size | 80 |
| 8.2 | Statistical Methods | 81 |
| 8.2.1 | Analysis Populations | 81 |
| 8.2.2 | Demographics and Baseline Characteristics | 81 |
| 8.2.3 | Primary Efficacy Endpoint(s) | |
| 8.2.4 | Secondary Efficacy Endpoint(s) | |
| 8.2.5 | Analysis of Safety | |

| Clinic | al Study . | Protoco | I: | BOS16172 | 1- | -02 |
|--------|------------|---------|----|----------|----|------|
| ъ. | 1.5 | 1 7 7 | | 2116 | 1 | 2016 |

| , |
|-------------------|

| 8.2.5.1 | Safety Analysis | 82 |
|---|---|---|
| 8.2.6 P | harmacokinetic and Pharmacodynamic Data | 82 |
| 8.2.6.1 | Analysis of Pharmacokinetic Data | 82 |
| 8.2.6.2 | Analysis of Pharmacodynamic Data | 83 |
| 8.2.6.3 | Population Pharmacokinetic Analysis or PK/PD Modeling | 83 |
| 8.3 Inter | m Analysis and Power | 83 |
| 9 ETHICS | S AND RESPONSIBILITIES | 83 |
| 9.1 Good | l Clinical Practice | 83 |
| | utional Review Board/Independent Ethics Committee | |
| 9.4 Infor | med Consent | 84 |
| | rds Management | |
| | ce Documentation | |
| | Files and Record Retention | |
| | ING AND MONITORING | |
| | OMENTS | |
| | REPORT AND PUBLICATIONS | |
| | DISCONTINUATION | |
| | DENTIALITY | |
| | ENCES | |
| | DICES | |
| APPENDIX | | |
| APPENDIX | | |
| APPENDIX | | |
| APPENDIX | | |
| APPENDIX | , | |
| APPENDIX<br>APPENDIX | | |
| ALLENDIA | LIST OF IN-TEXT TABLES | 101 |
| | DIST OF IN-TEXT TABLES | |
| Table 1. | Schedule of Assessments - Phase 1b - Multiple Ascending Dose | 42 |
| Table 2. | Schedule of Assessments - Phase 2 Proof of Concept (POC) Study | |
| Table 3. | Laboratory Tests | |
| Table 4. | Causality Definitions | 67 |
| | LIST OF IN-TEXT FIGURES | |
| Figure 1. | Individual pSTAT3 C <sub>min</sub> Levels Versus Dose | 28 |
| Figure 2. | Study Diagram for MAD Phase 1b and POC Phase 2 Studies | |

## LIST OF ABBREVIATIONS

ACR American College of Rheumatology

ADA anti-drug antibody
AE adverse event

AIDS acquired immune deficiency syndrome

ALT alanine aminotransferase
ANA antinuclear antibodies
ANC absolute neutrophil count
ANOVA analysis of variance
ANCOVA analysis of covariance
APL antiphospholipid

AST aspartate aminotransferase

AUC area under the concentration-time curve

AZA azathioprine

BICLA BILAG-based Composite Lupus Assessment

BILAG British Isles Lupus Assessment Group

BP blood pressure BUN blood urea nitrogen

BW body weight
C complement
CS corticosteroids

C-SSRS Columbia Suicide Severity Rating Scale

CD cluster of differentiation

CK creatine kinase C<sub>L</sub> systematic clearance

CLASI Cutaneous Lupus Erythematosus Area and Severity Index

C<sub>max</sub> maximum plasma concentration

CMH Cochran-Mantel-Haenszel

CS corticosteroids
CSR clinical study report
DILI drug-induced liver injury
DLT dose-limiting toxicity
DMC data monitoring committee

dsDNA double-stranded deoxyribonucleic acid

ECG electrocardiogram
EOT end of treatment

eCRF electronic case report form

F female

FAS full analysis set

CCI

BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02
Protocol Data and Varsion: 21 March 201


Fc fragment crystallizable

FDA Food and Drug Administration FSH follicle stimulating hormone

GCP Good Clinical Practice

eGFR estimated glomerular filtration rate

GLP Good Laboratory Practice

GWAS genome-wide association studies

γc gamma chain HBV hepatitis B virus

hCG human chorionic gonadotropin

HCl hydrochloride HCV hepatitis C virus

HIV human immunodeficiency virus

HR heart rate

HRT hormone replacement therapy

IA interim analysis

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonization

IEC Independent Ethics Committee

Ig immunoglobulin

IL interleukin

IL-21R interleukin 21 receptor

IM intramuscular INFy interferon gamma

INR International Normalized Ratio IRB Institutional Review Board

IUD intrauterine device

IV intravenous

IVRS interactive voice response system

JAK Janus kinase kg kilogram

KLH keyhole limpet hemocyanin LOCF last observation carried forward

M male

mAb monoclonal antibody
MAD multiple ascending dose

MAPK mitogen-activated protein kinase

MedDRA Medical Dictionary of Regulatory Activities

MS multiple sclerosis
MTX methotrexate

BOS161721 Boston Pharmaceuticals, Inc.


NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NIAID/FAAN National Institute of Allergy and Infectious Diseases/Food Allergy and

Anaphylaxis Network

NK natural killer

NOAEL no observed adverse event level

NO nitric oxide
OTC over-the-counter
PD pharmacodynamics
PEF peak expiratory flow

PGA Physician's Global Assessment

PK pharmacokinetics
POC proof of concept
PP per protocol

PR (interval) from onset of the p-wave to the end of the r-wave

pSS primary Sjögren's syndrome

pSTAT3 phosphorylated signal transducer and activator of transcription 3

PT preferred term

QRS (interval) from the onset of the q-wave to the end of the s-wave
QT (interval) from onset of the QRS complex to the end of the T wave
QTcF QT interval corrected for heart rate using Fridericia's formula

OFT-G QuantiFERON-TB Gold In-Tube

RA rheumatoid arthritis

RR (interval) from the onset of the r-wave to the onset of the next consecutive r-

wave

SAD single ascending dose SAE serious adverse event SAP statistical analysis plan

SC subcutaneous

SDMT safety data monitoring board

CCI

SLE systemic lupus erythematosus SLEDAI-2K SLE Disease Activity Index 2000

SLICC Systemic Lupus International Collaborating Clinics

Sm Smith

SOC system organ class
SRI-4 SLE Responder Index 4
SRI-5 SLE Responder Index 5
SRI-6 SLE Responder Index 6
SS safety analysis set

SSA Sjögren syndrome-A (Ro) SSB Sjögren syndrome-B (La) BOS161721 Boston Pharmaceuticals, Inc.


signal transducer and activator of transcription 3 STAT3

suspected unexpected serious adverse reaction **SUSAR** 

terminal elimination half-life  $t_{1/2}$ 

tuberculosis TΒ

T-cell dependent antibody response **TDAR** 

Tfh T-follicular helper

Th T-helper ΤK toxicokinetics

first time to maximum concentration  $T_{\text{max}}$ 

Treg regulatory T-cell TT tetanus toxoid

ULN upper limit of normal

**United States** US

volume of distribution Vd

WBC white blood cell

WHO World Health Organization WOCBP women of childbearing potential

triple mutation YTE

## 1. INTRODUCTION AND RATIONALE

#### 1.1 Indication

BOS161721 is a humanized monoclonal antibody (mAb), which binds to and inhibits interleukin-21 (IL-21) bioactivity, and is being developed for the treatment of moderately to severely active systemic lupus erythematosus (SLE) in adults.

## **1.2** Background and Rationale

#### 1.2.1 Overview of the Disease State

SLE is a chronic inflammatory autoimmune disease that has variable manifestations in multiple organ systems and follows a relapsing and remitting course. The disease process includes abnormal immune responses mediated by tissue-binding autoantibodies and immune complex deposition, giving rise to tissue damage often resulting in end organ disease and even mortality. Survival of SLE has improved due to earlier detection, improved overall medical care, and standardized SLE treatment with corticosteroids (CS), immunosuppressants, and cytotoxic agents. However, some of the morbidity in patients with SLE is related to its treatment. Comparison of early and late outcomes in patients with SLE demonstrate that death in early disease is most commonly due to infections and active SLE causing multi-system organ damage, while thromboses were the most common cause of death during later disease.

The reported prevalence of SLE in the United States (US) is 20 to 70 cases per 100,000 people. More than 90% of cases of SLE occur in women, frequently starting at childbearing age. Women of color are disproportionately affected by SLE. This suggests multiple genetic and environmental factors are at play. Accordingly, a multifactorial view of the immunopathogenesis of SLE suggests more than 1 area of interest, including breach in central tolerance in the adaptive arm of the immune system, peripheral amplification of the autoimmune response by the innate immune system, and local processes in the target organ that facilitate end-organ disease. 4

### **1.2.2 BOS161721 Development**

Boston Pharmaceuticals is developing BOS161721 for the treatment of SLE. BOS161721 is a humanized immunoglobulin G1 (IgG1) mAb directed against human IL-21.

Murine mAb 19E3, the progenitor of BOS161721, was generated using mouse hybridoma technology. 19E3 has subpicomolar (pM) affinity to human IL-21 and was selected for its potent neutralization of IL-21 bioactivity. BOS161721 was generated by the humanization of mAb 19E3 where its complementarity-determining regions were grafted onto a human IgG1 kappa backbone. The fragment crystallizable (Fc) portion of BOS161721 contains a YTE (M252Y/S254T/T256E triple mutation) in the constant domain of the IgG1 heavy chain that was introduced into the parental molecule, 19E3, intended to prolong the in vivo terminal elimination half-life (t<sub>1/2</sub>) of the mAb.<sup>5</sup> Thus, BOS161721 retains sub-pM binding to IL-21 and prevents IL-21 from binding to the IL-21 receptor (IL-21R), inhibiting IL-21 bioactivity.

BOS161721 binds to human IL-21 and Cynomolgus monkey IL-21, which are highly homologous, and neutralizes the bioactivity of both. BOS161721 is specific for IL-21 as it does not bind to or inhibit the other gamma-chain (γc) family of cytokines, and acts to specifically neutralize the IL-21 pathway. In *in vitro* studies, BOS161721 inhibited downstream IL-21-induced signaling, IL-21-induced plasma cell differentiation, and IL-21-induced natural killer (NK) cell activation. In *in vivo* studies, BOS161721 significantly inhibited the T-cell dependent antibody response (TDAR) to immunization with a protein antigen as well as B-cell expansion following a second protein antigen immunization in Cynomolgus monkeys.

#### **1.2.2.1 Interleukin-21**

IL-21 is an inflammatory cytokine, which belongs to a family of cytokines that also includes IL-2, IL-4, IL-7, IL-9, and IL-15, all of which bind to private receptors in complex with the common cytokine receptor yc. Most cytokines in this family are critically important for both the maintenance and function of T-cell and B-cell responses. IL-21 signals through a receptor complex consisting of its own private receptor, the IL-21R and vc. 6,7 Engagement of the IL-21R/γc complex leads to the activation of several signaling pathways, including the Janus kinase/signal transducer and activator of transcription, mitogen-activated protein kinase (MAPK) and phosphoinositide 3-kinase pathways. 8 IL-21 is produced mainly by T-cells and NK T-cells, but neutrophils have also been reported to produce IL-21. 9,10 The IL-21R is expressed on a broad array of cell types, including B-cells, T-cells, NK-cells, macrophages and dendritic cells, as well as other hematopoietic and nonhematopoietic cells such as fibroblasts, keratinocytes, and intestinal epithelial cells. 9,11 Activation of signal transducer and activator of transcription 3 (STAT3) via phosphorylation is critical in regulating human B-cell responses to IL-21<sup>12</sup>; phosphorylated STAT3 (pSTAT3) forms a homodimer, which translocates to the nucleus where it initiates transcription of the IL-21 gene, forming an autocrine loop for IL-21 production via STAT3 phosphorylation. <sup>13</sup> In addition, IL-21 has been shown to upregulate expression of its own receptor <sup>14</sup> and induces an autocrine feedback loop. <sup>15</sup>

IL-21 modulates various aspects of immune function. It promotes cluster of differentiation 4 (CD4+) T-cell differentiation and promotes the generation of T-helper (Th)17<sup>16</sup> and T-follicular helper (Tfh) cells. <sup>15,17</sup> In mice, IL-21 has been shown to regulate the balance between Th17 and regulatory T-cell (Treg), in that it increases Th17, while inhibiting Treg differentiation. <sup>18</sup> Less is understood with regards to human Tregs, although IL-21 has been reported to counteract Treg suppression of human effector T-cells and blockade of IL-21 promotes Treg generation in a murine model of graft versus host disease induced by human T-cells. <sup>20</sup> IL-21 upregulates CD8+ T-cell and NK-cell expansion and cytolytic activity by increasing granzyme B and perforin. <sup>21,22</sup> IL-21 also has been reported to increase granzyme B in plasmacytoid dendritic cells and B-cells resulting in inhibition of T-cell responses. <sup>23,24</sup> IL-21 also has a variety of effects on nonhematopoietic cells, such as stromal cells and induces inflammation through matrix metalloproteinase release by gut intestinal fibroblasts. <sup>25</sup>

One principal non-redundant role of IL-21 is the promotion of B-cell activation, differentiation, or death during humoral immune responses. <sup>14</sup> Furthermore, increased IL-21 production is characteristic of several autoimmune diseases and is likely to contribute to autoantibody production as well as pathologic features of autoimmune disease. <sup>26</sup> The critical role of IL-21 in promoting humoral and other immune responses makes it an important focus of potential

therapeutic interventions in conditions characterized by overproduction of pathogenic autoantibodies. IL-21 production by Tfh cells in humans is believed to play a major role in driving the autoantibody production through its role in plasma cell differentiation. Importantly, Tfh cell populations are expanded in patients with autoimmune diseases such as lupus, bullous pemphigoid, rheumatoid arthritis (RA) and primary Sjögren's syndrome (pSS) and have been reported to correlate with IL-21 levels, autoantibodies, and disease severity. <sup>26,27,28,29</sup> Furthermore, loss of number and functionality of Tregs has been associated with autoimmune diseases such as SLE and giant cell arteritis, which IL-21 is expected to modulate. <sup>30,31</sup> Thus, neutralization of IL-21 in settings of autoimmunity is expected to impact several cell populations believed to be involved in the pathogenesis of autoimmune disorders including SLE.

BOS161721 selectively binds IL-21 with high affinity to neutralize IL-21, and due to its pleiotropic nature, neutralization of IL-21 is expected to impact several cell populations believed to be involved in the pathogenesis of SLE. Importantly, patients with SLE have elevated IL-21 plasma levels that correlate with the severity of the disease. Recently, genome-wide association studies (GWAS) have provided convincing evidence that the chromosomal 4q 27 region harbors the IL-21 genes and is associated with chronic inflammatory disorders, including SLE.<sup>29</sup>

#### 1.2.2.2 Preclinical Studies

The pharmacokinetics (PK) of BOS161721 were characterized following single-dose intravenous (IV) administration of BOS161721 (0.01 to 30 mg/kg) in male Cynomolgus monkeys or repeat, every 2 weeks IV administration (15 to 100 mg/kg) and subcutaneous (SC) administration (50 mg/kg) in male and female Cynomolgus monkeys. Systemic exposure was approximately dose-proportional within the tested dose range. SC bioavailability was determined to be 64.3%.

Two single-dose (IV) non-good laboratory practice (GLP) studies conducted in Cynomolgus monkeys evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), and immunogenicity of BOS161721. Following a single IV administration (slow bolus), there were no BOS161721-related adverse changes, resulting in a no-observed-adverse-effect-level (NOAEL) value of 30 mg/kg, the highest dose tested among 2 studies.

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) administration for 3 months (a total of 7 doses).



## 1.2.2.3 Clinical Studies

BOS161721-01 was a double-blind, Phase 1, single ascending dose (SAD) study to assess the safety, PK, and PD of BOS161721 in healthy subjects. The primary objective of the study was to characterize the safety and tolerability of IV and SC SADs of BOS161721 in an otherwise healthy subject population without concomitant illnesses, immune abnormalities, or concomitant medications. Secondary objectives included characterization of the PK and immunogenicity of BOS161721, and exploratory objectives included the evaluation of the effect of BOS161721 on TDAR to keyhole limpet hemocyanin (KLH) (primary and secondary immunizations) in healthy subjects, the effects of BOS161721 on plasma levels of IL-21 (free and bound), and the evaluation of the effect of BOS161721 on IL-21 gene expression (via gene signature) in blood. This study consisted of 8 cohorts. Subjects were randomized in a 3:1 ratio (BOS161721: placebo) and received either a single dose of BOS161721 (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) or placebo, with safety follow-up. For the first cohort, after the first 2 subjects were dosed (1 active and 1 placebo), there was a minimum gap of 48 hours before the remaining subjects from that cohort were dosed, to allow for an initial review of any emerging safety and tolerability data. For all cohorts, escalation to the next dose was not sooner than 8 days after all the subjects in the prior cohort had been dosed and were based on a review of at least 7 days of safety and tolerability data by the Safety Data Monitoring Team (SDMT).

Blood samples were collected at every in-house study visit for BOS161721 concentration determinations. Blood samples were also collected for determination of IL-21 plasma levels (free and total). Safety was assessed based on the occurrence of treatment-emergent AEs, hepatic function abnormality, and acute and delayed hypersensitivity reactions. Other safety variables included electrocardiograms (ECGs), vital signs (blood pressure [BP], heart rate, and temperature), safety laboratory assessments, blood sampling for ADAs, total IgG and immunoglobulin M (IgM) levels, CD4+ count, and full and targeted physical examinations. Overall, there were no clinically significant findings from this study, following an interim cut and review of the data at Day 90 postdose. Adverse events reported as related to the study drug, particularly infections, were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. There was 1 serious adverse event (SAE; death due to pulmonary embolism) that occurred 127 days after a single administration of 240 mg SC dose of BOS161721. The causality of this single SAE was not attributed to study drug and further information can be found in the Investigator's Brochure. PK data from the SAD study demonstrates BOS161721 has an extended  $t_{1/2}$  (provisional single dose data indicates this to be approximately 42-46 days) which supports evaluation of monthly dosing.

## 1.2.3 Study Dose Selection

Doses have been selected for the multiple ascending dose (MAD) Phase 1 study based on a 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01); the SDMT reviewed the blinded safety data from subjects for each dose cohort (8 cohorts, evaluating 1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg), along with the accumulated safety and available PK/PD data from all subjects in the previous dose cohorts, to make a decision on whether to proceed to the next higher dose level, repeat a dose level, or stop dose escalation. Overall, there were no clinically significant safety or tolerability findings from this study.

Based on the Day-90 interim cut of the PK and biomarker data in the BOS161721-01 study, the recommended doses for evaluation in the MAD phase of this study are 20, 60, and 120 mg SC monthly. This dose recommendation is supported by evidence of linear PK with BOS161721 resulting in a median first time to maximum concentration (T<sub>max</sub>) of 6 days and an apparent terminal half-life of 44 days. Furthermore, pSTAT3 suppression, a marker of IL-21 target engagement, follows a similar time course of the mAb levels, with maximal and sustained suppression apparent with doses greater than 30 mg SC (Figure 1).



Figure 1. Individual pSTAT3 C<sub>min</sub> Levels Versus Dose

IV = intravenous, pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SC = subcutaneous

All doses selected for the MAD study are projected not to exceed the mean exposure of that achieved following the highest single dose of 240 mg SC administered in the Phase 1 SAD study. Cohort 1 will include randomized treatment to the 20 mg dose. Based on the staggered study design, the data monitoring committee (DMC) will perform a scheduled review of safety data and sequentially consider dose escalation for Cohorts 2 and 3. In addition, the DMC and Boston Pharmaceuticals will conduct a data review to suggest which dose should be carried forward into the proof of concept (POC) Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD study (see Section 3.1.1.1).

#### 1.2.4 Risk-Benefit Assessment

The available preclinical data on BOS161721, the findings in clinical study BOS161721-01, and existing clinical information on IL-21 inhibitors suggest that the present clinical study has an acceptable risk-benefit ratio. In this study, the risk-benefit assessment of BOS161721 in adult patients with moderately to severely active SLE will be ongoing, with step-wise evaluations during the staggered MAD study. The DMC used in this study is charged with assessing such actions in light of an acceptable benefit-risk profile for BOS161721 as an anti-IL-21 mAb. Formal DMC monitoring meetings will occur as described in the DMC Charter. Two weeks after Cohort 1 has received a second dose of study drug, the DMC will evaluate the safety and tolerability data from Cohort 1 to determine the recommended dose for Cohort 2. Two weeks after 8 patients in Cohort 2 receive a second dose, the DMC will determine if dose escalation to Cohort 3 can proceed. Two weeks after the last patient in Cohort 3 receives the second dose, the DMC and Boston Pharmaceuticals will conduct a data review to suggest which dose should be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 during the MAD study. Thereafter, DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter. With the agreement of the DMC and sponsor, this schedule may be modified depending on the rate of patient accrual. Additional details can be found in the DMC Charter.

The benefit of participation for all patients in this study is close monitoring of their medical condition and safety of their treatment. Those randomized to the active treatment arm may potentially experience improvement in their SLE disease. Those randomized to the placebo (in combination with standard of care) arm are not expected to obtain any additional benefit, beyond those of their background treatment, though close monitoring of their medical condition and safety may itself be associated with improving their SLE.

#### 1.2.5 Potential Risks

Potential risks based on the mechanism of action of BOS161721 include infections, risks associated with the administration of any foreign protein or biologic agent, including injection site reaction, anaphylaxis, serious allergic reaction, and development of ADAs. ADAs could result in immune complex disease (with manifestations such as arthralgias, serum-sickness, and vasculitis), autoimmunity, or altered BOS161721 levels or activity. Further details can be found

in the current Investigator's Brochure (IB) for BOS161721, which contains comprehensive toxicology, preclinical and clinical information on BOS161721.

Two investigational drug products are considered to be in the same pharmacological class as BOS161721 based on interruption of signaling through the IL-21 signaling pathway. No potential risk generalizable across the class has been observed with these investigational products. Based on the clinical Phase 1 SAD study (BOS161721-01), AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs.

The majority of IgG elimination occurs via intracellular catabolism, following fluid-phase or receptor-mediated endocytosis. This type of endocytosis and elimination is a form of target-mediated disposition where the interaction of the drug and its pharmacological target (eg, a target receptor) serves as a significant contributor to the kinetics of antibody distribution and elimination. Renal elimination, which is a primary pathway of clearance of small-molecule drugs, is relatively unimportant for IgG, as its large size prevents efficient filtration through the glomerulus. Secretion into the bile is an important pathway of elimination of IgA antibodies, but this route is not a significant contributor to the elimination of IgG antibodies. Thus, risk to renal and hepatic systems due to metabolism of BOS161721 is low.<sup>33</sup>

## 1.2.5.1 Anaphylaxis and Serious Allergic Reactions

As with the administration of any foreign protein and/or other biological agents, acute hypersensitivity reactions, including acute anaphylactic/hypersensitivity, severe allergic, and anaphylactoid reactions may follow infusion of mAbs and can be caused by various mechanisms. These acute hypersensitivity reactions may be severe and result in death.

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria,<sup>34</sup> and are discussed in Section 6.2.2.6.1.

Based on the limited Phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed.

Patients with a known history of allergy or severe hypersensitivity reaction to any component of BOS161721 formulation or patients with a history of anaphylaxis to any other biological therapy such as mAbs will be excluded from studies with BOS161721. In addition, appropriate drugs and medical equipment to treat acute hypotensive, bronchoconstrictive, or anaphylactic reactions will be immediately available at the unit and study personnel will be trained to recognize and treat these reactions.

#### 1.2.5.2 Injection Site Reactions

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) for 3 months (a total of 7 doses); no SC animals had injection reactions.

Based on the Phase 1 SAD study (BOS161721-01), incidence of injection site reactions in subjects who received BOS161721 was similar to placebo.

Patients will be monitored for local injection site reactions in this study. See Section 6.2.7.

## **1.2.5.3 Immune Complex Disease**

The potential risk of immune complex disease for BOS161721 is theoretical, based on the known risks associated with mAbs. The administration of a mAb can result in the formation of ADAs. Administration of the mAb in the presence of ADA may result in the formation of circulating antibody-antigen complexes potentially resulting in altered BOS161721 levels or activity or deposition of the complexes in microvasculature. Complement is frequently involved in the latter setting, and the breakdown products of complement attract polymorphonuclear leukocytes to the site of deposition where they can provoke local tissue damage through specific or nonspecific release of enzymes. Two of the more common end-organ targets are the blood vessels (vasculitis) and kidney (nephritis). These clinical manifestations represent immune complex disease or Type III hypersensitivity. Although BOS161721 is a humanized mAb, ADAs may develop; however, the likelihood of occurrence of immune complex disease with BOS161721 is low. The findings of immune complex disease are typically reversible when mAb administration stops and the antibody-antigen complexes are cleared from the body.

Based on the limited Phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed.

#### 1.2.5.4 Infections

BOS161721 is expected to diminish the activity of T-cell, B-cell and NK-cell lines. Like other medications modulating immune response, BOS161721 may increase the potential risk for infection, including serious infections. IL-21 produced by CD4+ Th cells is required to sustain the anti-viral function of CD8+ T-cells against chronic viral infections. Nonclinical evidence suggests that the risk of chronic viral infection recurrence or increased severity may occur with IL-21 inhibition.<sup>35</sup>

These conditions will be fully characterized with clinical descriptions and routine laboratory and/or specialty testing and treated where indicated with appropriate local standard of care.

Patients with a history of opportunistic infection, including recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years, or any other underlying pathology predisposing to serious infection, are excluded from studies with BOS161721 (for further details please refer to the current IB for BOS161721).

Patients will be assessed for hepatitis B, and C, and HIV-1/2 combination, at screening.

## Cryptosporidium Infection

Cryptosporidium infection was noted in patients with an IL-21 receptor loss-of-function gene mutation and similar findings of cryptosporidium infection have been observed in immunosuppressed liver transplant and human immunodeficiency virus patients. <sup>36,37</sup> Since
BOS161721 is expected to diminish the immunosurveillance activity of T-cell, B-cell, and NK-cell lines, a similar risk is biologically plausible with prolonged exposure to BOS161721.

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells,<sup>37</sup> patients with a CD4+ count < 500 cell/mm<sup>3</sup> were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from the proposed MAD/POC studies. Patients exposed to investigational product who develop diarrhea during the course of the study should immediately undergo an assessment for opportunistic infection including stool for ova and parasites and stool examination for cryptosporidium. Positive cryptosporidium in stool sample at screening is an exclusion. Treatment by the investigator where indicated should be guided by findings and be consistent with local standard of care.

Based on the limited Phase 1 SAD study (BOS161721-01), infections in subjects who received BOS161721 was not observed.

# 1.2.5.5 Malignancy

The stimulatory effect of IL-21 on NK cells and CD8+ T-cells suggests the cytokine may have anti-tumor activity. Nonclinical studies have demonstrated significant anti-tumor effects of IL-21 in a number of tumor models. IL-21 therapy of human metastatic melanoma and renal cell carcinoma has demonstrated POC with significant increases in levels of perforin, granzyme B, and interferon gamma (IFN $\gamma$ ) expression in CD8+ T-cells and NK T-cells. Clinical response has been limited in these generally unmanageable diseases.

The impact of treatment with anti-IL-21 therapy on the development or growth of malignancies is not known; however, as with other immunomodulatory biologic agents, treatment with BOS161721 may result in an increase in the risk of malignancies. NK cell suppression by IL-21 neutralization may represent a biological mechanism for a potential risk for malignancy. Patients with a history or current diagnosis of cancer within the past 5 years, with the exception of non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy, are excluded from the study.

Based on the limited Phase 1 SAD study (BOS161721-01), malignancy in subjects who received BOS161721 was not observed.

## **1.2.5.6** Hepatic Function Abnormality

There is no substantial evidence suggesting BOS161721 is associated with liver function abnormality. However, as a precaution, patients with a history of abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST >  $2 \times \text{upper limit of normal [ULN]}$ ; total bilirubin >  $1.5 \times \text{[ULN]}$  and judged by the investigator to be clinically significant) were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from the MAD study. Patients with a positive hepatitis B or C test or a history of alcohol dependence will also be excluded.

Based on the limited Phase 1 SAD study (BOS161721-01), hepatic function abnormality in subjects who received BOS161721 was not observed.

### 1.2.5.7 Failure of Vaccination

IL-21 is a key cytokine in development of B-cells into immunoglobulin-secreting plasma cells. Abnormal signaling through the IL-21R/Janus Kinase (JAK)3/signal transducer and activator of transcription (STAT3) pathway leads to defective humoral immune responses to both T-dependent and T-independent antigens and impairs the establishment of long-lasting B-cell memory. Abnormal signaling through the pathway has been related to decreased specific antibody responses following vaccination, and to increased susceptibility to encapsulated bacterial infections.<sup>38</sup>

The effect of BOS161721 was evaluated in in vivo single dose studies in Cynomolgus monkey in which the animals received vaccination to T-cell dependent KLH antigen to stimulate a TDAR. These in vivo studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen; however, it is worth noting that BOS161721 administration did not produce any remarkable changes in anti-KLH antibody data for IgM, IgG1, IgG3, and IgG4 or anti-tetanus toxoid (TT) antibody data for IgM, IgG, IgG1, or IgE during the dosing phase in the same study.

# 1.2.5.8 Potential for Drug-Drug Interactions

Drug-drug interactions were not evaluated in the Phase 1 SAD study (BOS161721-01), which included only healthy adult subjects. Use of prescription medications (with the exceptions of oral contraceptives), and over-the-counter (OTC) treatments including herbal supplements such as St John's Wort (except multivitamins), in the 2 weeks prior to screening was prohibited in the SAD study.

See Section 4.5 for other specific exclusion criteria which support lowered risk of interactions, and Section 4.6.1 for corticosteroid (CS) dosing. In addition, Section 1.2.5.6 describes considerations for hepatic function for this study.

## 1.2.5.9 Potential Risk to Fetal Development

No data on preclinical reproductive toxicity are available at the time of this study.

# 2 STUDY OBJECTIVES AND ENDPOINTS

This trial has separate objectives and endpoints for the MAD Phase 1b and POC Phase 2 studies. The primary, secondary, and exploratory objectives for each phase, as applicable, are described below with their corresponding endpoints.

# 2.1 Phase 1b Multiple Ascending Dose

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose. | <ul> <li>Safety Endpoints</li> <li>Incidence and severity of AEs and SAEs, related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness</li> <li>Injection site reactions</li> <li>Columbia Suicide severity Rating Scale (C-SSRS)</li> <li>12-lead ECGs parameter results at each visit and change from baseline</li> <li>Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline</li> <li>Clinical laboratory results and change from baseline</li> <li>Physical examinations changes from baseline</li> <li>ADAs</li> <li>Study drug exposure/compliance</li> <li>Concomitant medication usage</li> </ul> |
| Secondary | concentiant incurrence usage |
| To characterize the PK of BOS161721 and select the optimal dose of BOS161721 based on safety, PK, and PD effects in patients with mild to moderate SLE. | <ul> <li>Pharmacokinetic Endpoints</li> <li>BOS161721 concentration by visit and time point</li> <li>Maximum observed concentration (C<sub>max</sub>), T<sub>max</sub>, area under the concentration-time curve (AUC), terminal elimination half-life (t<sub>½</sub>), systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>)</li> <li>Pharmacodynamic Endpoints</li> <li>Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype</li> <li>Results and changes (or shifts) from baseline in antidouble-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit</li> <li>Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit</li> </ul> |



# 2.2 Phase 2 Proof of Concept

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To demonstrate a superior effect of<br>BOS161721 at the chosen dose compared<br>with placebo for response on the SRI-4 | Primary Efficacy Endpoint The proportion of subjects with a SRI-4 response at Day 210 (see Section 6.3.4.1) |
| Secondary | |
| To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult | Secondary Efficacy Endpoints The proportion of subjects with: SRI-4 response at each visit |

patients with moderately to severely active SLE on limited background standard of care treatment

- SRI-5 and SRI-6 response (Section 6.3.4.2)
- a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210
- new BILAG A flare or > 1 BILAG B flares relative to baseline through Day 210
- PGA worsening
- a BICLA response
- a CLASI response
- medication failures
- Results and changes from baseline in:
  - CLASI
  - swollen and tender joints ACR-28
  - SLEDAI-2K
  - SLICC/ACR damage index
  - Time to medication failure
- Duration of SRI-4 response
- Time to first SRI-4 response
- Time to BILAG A flare or > 1 BILAG B flare compared to baseline through Day 210

### Safety

 To assess safety and tolerability of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment

#### Safety Endpoints

- Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness
- Injection site reactions
- C-SSRS
- 12-lead ECGs parameter results at each visit and change from baseline
- Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline
- Clinical laboratory results and change from baseline
- Physical examinations changes from baseline
- ADAs
- Study drug exposure/compliance
- Concomitant medication usage

#### **Exploratory**







## 3 STUDY PLAN

# 3.1 Study Design

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly.

The trial will consist of 2 double-blinded studies: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.

SLE disease activity assessment data will be centrally reviewed by medical monitor and sponsor to ensure the scores are clinically meaningful and compliant with specific definition. The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease being studied. Further details on the content and methods of data reports by the medical monitor and sponsor will be outlined in the Medical Data Review Plan along with the processes and procedures that will be followed.

## 3.1.1 Multiple Ascending Dose Phase 1b Study

The MAD study will consist of 3 cohorts:

- Cohort 1 (20 mg SC) will include 6 patients
  - 5 patients will receive BOS161721 (active group) and 1 patient will receive placebo (placebo group)
- Cohorts 2 (60 mg SC) and 3 (120 mg SC) will include 12 patients each
  - o 9 patients in the active group and 3 in the placebo group

Doses selected for each of the 3 cohorts is based on a 90-day safety, tolerability, PK and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. All doses selected for

the MAD study are projected not to exceed the mean exposure of that achieved in the SAD study.

## 3.1.1.1 Dose Escalation for the MAD Study

The MAD study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after DMC evaluation of the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after DMC evaluation of the safety and tolerability data from Cohorts 1 and 2. Each cohort will continue at their assigned dose level through their respective 6-month treatment periods (See Study Schematic, Section 3.1). If patients discontinue the study in a cohort prior to adequate safety follow-up, he/she may be replaced.

Criteria for dose escalation are further described in the DMC Charter. See Section 3.1.1.2 for additional details about DLTs.

## 3.1.1.2 Dose Limiting Toxicity (DLT)

Severity of adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs occurring after study drug administration, which are attributable to the study drug, will be considered DLTs:

## **Hematologic:**

- Grade 4 neutropenia
- Grade 3 neutropenic infection
- Grade 3 thrombocytopenia with bleeding
- Grade 4 thrombocytopenia

### **Non-Hematologic:**

- Grade 3 or above toxicities, persisting after optimal treatment with standard medical therapy (eg, anti-emetics, anti-diarrheals)
- Drug-induced liver injury ([DILI], Hy's Law), as defined in Section 6.2.2.6.3

Investigators should always manage their patients according to their medical judgment which may include interruption of study drug based on the particular clinical circumstances.

## 3.1.1.3 DMC Recommendations

During scheduled meetings, the DMC will review relevant study data for safety or benefit-risk concern. During the MAD study, the DMC may provide the following recommendations to the sponsor:

- Expanding a cohort at a specific dosing level, or repeating a lower dose in a subsequent cohort
- Continuing a dose level for a given cohort
- Escalating a dose level for a subsequent cohort
- Termination of current or previous cohort(s)

Further dosing in a given cohort will be halted if 2 or more DLTs are identified intra- and inter-patients dosed. For the POC study, the DMC and Boston Pharmaceuticals will conduct a data review to suggest which dose should be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available at the time the last patient in Cohort 3 completes the Day 44 visit (2 weeks after dose 2). Details are provided in the DMC Charter.

# 3.1.2 POC Phase 2 Study

### 3.1.2.1 BOS161721 Dose

The optimal dose evaluation is chosen based on MAD Phase 1b safety, tolerability, immunogenicity, and PK and PD data. The dose will be communicated by a letter to site investigators participating in the POC Phase 2 study, and to the IRB/IEC.

# 3.1.2.2 POC Study Design

For the POC study, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio.

As in the MAD study, each patient in the POC study may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Section 3.4). Dose selection will be based on the DMC and sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD study of 30 patients treated with BOS161721/placebo.

DMC safety reviews will be conducted periodically throughout the study as described in the DMC charter.

# 3.2 Randomization and Blinding

This is a randomized, double-blind study.

Patients meeting all inclusion and exclusion criteria will be centrally randomized to either placebo or BOS161721 using an IWRS according to a randomization list generated by an independent, non-study statistician. Randomization will be performed separately for each study phase and separately for each cohort in the Phase 1b and 2 portions as follows:

| Phase/Cohort | Number of Patients | Randomization Ratio BOS161721:Placebo |
|---|---|---|
| Phase 1b/Cohort 1 | 6 | 5:1 |
| Phase 1b/Cohort 2 | 12 | 3:1 |
| Phase 1b/Cohort 3 | 12 | 3:1 |
| Phase 2 | 156* | 2:1 |

<sup>\*</sup>Additional patients may be enrolled to confirm sufficient numbers of patients are in the full analysis set (FAS).

Eligible patients will be assigned to the study phase which is active at time of enrollment. Similarly, patients in the Phase 1 MAD will be assigned to the cohort which is active. Each patient will be assigned a unique randomization number which will not be reused.

All patients, investigators, and study team participants will be blinded to treatment assignment. An independent biostatistician not otherwise involved on the study will be unblinded and prepare materials for the interim analysis (IA) and the DMC safety reviews. The DMC will review unblinded data during safety reviews and the IA. A limited team at Boston Pharmaceuticals will review unblinded results from the Phase 1b MAD portion during the IA to determine the dose that will be used for the Phase 2 POC portion of the study. Details regarding maintenance of the blinding and content of data reviews will be described in the DMC charter or related study documentation.


# 3.3 Study Schematic

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2 Studies



A = active drug (BOS161721); P = placebo


# 3.4 Schedule of Assessments

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen | Enroll | | | | | | | | | | | | Safet | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | - | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | - | 11 | 12 | 13 |
| GENERAL ASSESS | MENTS | | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| SLICC Criteria for<br>SLE | X | | | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>c</sup> | | X | | | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | | X | | X | X | X | X | X | | | | | |
| SAFETY ASSESSM | ENTS | | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | | | |
| Chest x-ray <sup>d</sup> | X | | | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>e</sup> | X | X | | | X | | | X | | | | | | | | X |
| Injection site reaction assessment | | X <sup>f</sup> | X | | X | | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | | X | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>g</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESS | SMENTS | | | | | | | | | | | | | | | |
| BILAG-2004 Index | X | X | | | X | | X | X | X | X | X | | | X | X | X |


Schedule of Assessments - Phase 1b - Multiple Ascending Dose Table 1.

| | Screena | Enroll | | | | Tre | eatment | Period | Follow- | Up | | | | Safet | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| SLEDAI-2K | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| PGA of disease activity | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CCI | 71 | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLICC/ACR<br>Damage Index | | X | | | | | | | | | X | | | | | |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| LABORATORY ASS | SESSMEN | l | | | | | | | | | | | | | | 111 |
| CD4+ count | X | X | | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments (hematology and | | | | | | | | | | | | | | | | |
| clinical chemistry) <sup>h</sup> | X | X | | | X | X | X | X | X | X | X | | | X | X | X |
| Coomb's test direct <sup>i</sup> | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | | X | X | X | | X | | | X | | | | | |
| Plasma CCI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Plasma CCI & | | X | | X | X | | X | X | | | X | | | | | |
| Whole blood for leukocyte | | | | | | | | | | | | | | | | |
| immunophenotype | | X | | X | X | | X | X | | | X | | | | | |
| ADA <sup>j</sup> | | X | | X | X | | X | X | | | X | | | | | X |
| nAb <sup>k</sup> | | | | | | | | X | | | X | | | | | |
| pSTAT3 <sup>1</sup> | | X | | | X | X | X | X | | | | | | | | |
| CCI | | X | | X | | | | X | | | X | | | | | X |
| CCI | | X | | | | | | | | | | | | | | ] |


Schedule of Assessments - Phase 1b - Multiple Ascending Dose Table 1.

| | Screena | Enroll | | | | | | | | | | | Safet | y Follow | v-Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| CCI | X | X | | | X | | X | X | X | X | X | | | X <sup>m</sup> | X <sup>m</sup> | X <sup>m</sup> |
| CRP | X | | | | | | | X | | | | | | | | X |
| Serum pregnancy<br>test (women) | X | | | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>n</sup> | | X | | | X | | X | X | X | X | X | | | | | |
| TB test<br>(QuantiFERON-TB<br>Gold In-Tube) <sup>d</sup> | X | | | | | | | | | | | | | | | |
| Serology (hepatitis<br>B and C, HIV-1/2<br>combination) | X | | | | | | | | | | | | | | | |
| Stool sample <sup>o</sup> | X | | | | | | | | | | | | | | | |
| Spot urine for protein/creatinine ratio | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | | X | | X | X | X | X | X | | | X X X | | |
| PK Labs | | | | l | | l | | | | <u> </u> | l | | l | | l | |
| Predose | | X | | | X | | X | X | X | X | X | | | | | |
| Postdose | | X <sup>q</sup> | X | X | X <sup>q</sup> | | | | | | X <sup>q</sup> | X | X | X | X | X |


Clinical Study Protocol: BOS161721-02


 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | Tre | atment | Period | Follow- | Up | | | Safet | Safety Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 30 44 60 90 120 150 180 187 19 | | | | | | 195 | 210 | 240 | 270 | |
| Days | to -1 | 0 | (± 1) | | | | | | | | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 4 5 6 7 8 9 10 | | | | | | | 11 | 12 | 13 | |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CCl ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CCl

; FSH = follicle stimulating hormone; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G;

IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; nAb = neutralizing antibody; PGA = Physician's Global Assessment;

PK = pharmacokinetic; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SAE = serious adverse event; SC = subcutaneous; CCI

; SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; TB = tuberculosis; TDAR = T-cell dependent antigen response.

<sup>a</sup> Screening assessments will be performed over more than 1 visit.

- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 4.6.1 for further details.
- c Randomization should occur after patient eligibility has been confirmed by central eligibility review.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- <sup>e</sup> ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed at 2 hours postdose.
- Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, 187, and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.
- h Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.
- When clinically indicated for hemolytic anemia.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.
- <sup>k</sup> nAb is assessed if patient is positive for ADA.
- Predose (trough) samples only.
- <sup>m</sup> Only dsDNA collected during safety follow-up visits.
- <sup>n</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- Oryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- Postdose samples will be collected at 4, 8, and 24 hours after study drug administration on Days 0, 30, and 180.


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screen <sup>a</sup> | Enroll Treatment Period Follow-up | | | | | | | | | | Safe | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| GENERAL ASSESSMENTS | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| SLICC Criteria for SLE | X | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>c</sup> | | X | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | X | X | X | X | X | X | | | | | |
| SAFETY ASSESSMENTS | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | |
| Chest x-ray <sup>d</sup> | X | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>e</sup> | X | X | | X | | X | | | | | | | | X |
| Injection site reaction assessment | | $X^{f}$ | | X | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>g</sup> | X | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESSMENTS | ľ | 1 | | | | I. | I. | I. | | | I. | l . | II. | |
| BILAG-2004 Index | X | X | | X | X | X | X | X | X | | | X | X | X |
| SLEDAI-2K | X | X | | X | X | X | X | X | X | | | X | X | X |
| PGA | X | X | | X | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | X | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | X | X | X | X | X | X | | | X | X | X |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screena | een <sup>a</sup> Enroll Treatment Period Follow-up | | | | | | | | | Safe | ty Follo | w_Un | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | Emon | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| SLICC/ACR Damage Index | | X | | | | | | | X | | | | | |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |
| LABORATORY ASSESSMENT | ΓS | | | | | | | | | | | | | |
| CD4+ count | X | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments (hematology and clinical | V | 37 | | | 37 | 37 | 37 | | 37 | | | | 37 | 37 |
| chemistry) <sup>h</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Coomb's test direct | X | X | 37 | | X | | X | X | | | | X | X | X |
| Total IgG and IgM | X | X | X | X | 37 | X | 37 | 37 | X | | | 37 | 37 | 37 |
| Plasma CCI | X | X | 37 | X | X | X | X | X | X | | | X | X | X |
| Plasma CCI & CCI | | X | X | X | | X | | | X | | | | | |
| Whole blood for leukocyte immunophenotype | | X | X | X | | X | | | X | | | | | |
| ADA <sup>j</sup> | | X | X | X | X | X | | | X | | | | | X |
| nAb <sup>k</sup> | | | | | | X | | | X | | | | | |
| CCI | | X | X | | | X | | | X | | | | | X |
| CCI | | X | | | | | | | | | | | | |
| CCI | X | X | | X | X | X | X | X | X | | | X <sup>l</sup> | X <sup>l</sup> | X <sup>l</sup> |
| CRP | X | | | | | X | | | | | | | | X |
| Serum pregnancy test (women) | X | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>m</sup> | | X | | X | X | X | X | X | X | | | | | |
| TB test (QuantiFERON-TB<br>Gold In-Tube) <sup>d</sup> | X | | | | | | | | | | | | | |
| Serology (hepatitis B and C,<br>HIV-1/2 combination) | X | | | | | | | | | | | | | |
| Stool sample <sup>n</sup> | X | | | | _ | | | | | | | | | |


Clinical Study Protocol: BOS161721-02


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screena | Enroll | | | Tı | eatment | Period 1 | Follow-u | p | | | Safe | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | $(\pm 3)$ | (± 3) | $(\pm 3)$ | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | $(\pm 3)$ | (± 3) | (± 3) | $(\pm 3)$ |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | - | | 10 | 11 | 12 |
| Spot urine for protein/creatinine | | | | | | | | | | | | | | |
| ratio | X | X | | X | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | X | X | X | X | X | X | | | X | X | X |
| PK Labs <sup>o</sup> | | | | | | | | | | | | | | |
| Predose | | X | | X | X | X | X | X | X | | | | | |
| Postdose | | | X | | | | | | | X | X | X | X | X |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CCl ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CCl ; FSH = follicle stimulating hormone; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; SAE = serious adverse event; SC = subcutaneous; CCl ; SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; CCl dependent antigen response.

- <sup>a</sup> Screening assessments will be performed over more than 1 visit.
- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 4.6.1 for further details.
- Randomization should occur after patient eligibility has been confirmed. The actual randomization procedure can be completed on Day -1 after eligibility confirmation or the morning of Day 0 prior to dosing for logistical purposes.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- <sup>e</sup> ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed at 2 hours postdose.
- Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 187 and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.
- h Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.
- When clinically indicated for hemolytic anemia.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.


Clinical Study Protocol: BOS161721-02


Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screena | Enroll | | | Tı | reatment | Period 1 | Follow-u | p | | | Safe | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 4 5 6 7 8 9 10 11 12 | | | | | | | | | | | |

half is assessed if patient is positive for ADA.


Only CCI collected during safety follow-up visits.

<sup>&</sup>lt;sup>m</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.

<sup>&</sup>lt;sup>n</sup> Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

<sup>&</sup>lt;sup>o</sup> PK samples will only be collected at the investigational sites that will be participating in the PK portion of the study.

## 4 POPULATION

# 4.1 Participant Recruitment

Advertisements approved by the IRB, and investigator databases, may be used as recruitment procedures for adult men and women with moderately to severely active SLE.

#### 4.2 Number of Patients

Approximately 186 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD Phase 1b study, and approximately 156 additional patients will be randomized in the POC Phase 2 study. Note that approximately 24 dropouts are assumed.

# 4.3 Patient Screening

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Section 3.4]) for this study must be performed between Day -28 and Day -1.

## 4.4 Inclusion Criteria

Patients who meet the following criteria will be considered eligible to participate in this clinical study:

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion or Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
  - c. C3 or C4 below normal as determined by central lab

Clinical Study Protocol: BOS161721-02


- 5. At screening, the SLE Disease Activity Index 2000 (SLEDAI-2K) must be ≥ 6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 7. Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - i. "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis in ≥ 2 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living that has been present on several days cumulatively over the past 30 days, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
      - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):
        - Ambulation, toileting, grooming- including bathing and dressing; feeding oneself
    - ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in ≥ 1 joint, (observed or throughout history), with some loss of functional range of movements which lead to some loss of functional range of motion as manifested by effects on instrumental ADLs such as:

• Cooking, driving, using the telephone or computer, shopping, cleaning, etc, and has been present on several days over the last 30 days, and is present at the time of the screening visit

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization) (see APPENDIX 3)
- 9. Women of childbearing potential (WOCBP; see Section 4.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

### 4.5 Exclusion Criteria

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study


- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed.
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study. (See Section 4.6 for prohibited concomitant medication)
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count < 500/μL at screening
- 16. Platelets < 50,000/mm $^3$  (50  $\times$  10 $^9$ /L) or < 35,000/ mm $^3$  (35  $\times$  10 $^9$ /L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if due to anemia related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)

19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation <sup>39</sup>:

- GFR = ([1 for male] or [0.85 for female])  $\times$  (140 Age)  $\times$  BW / (72  $\times$  Creatinine)
- 20. Serum ALT and/or serum AST > 2  $\times$  ULN at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK)  $> 3.0 \times$  ULN at screening, unless it is related to lupus myositis
- 22. Direct bilirubin  $> 1.5 \times ULN$  at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (eg, IgG protein) or molecules made of components of monoclonal antibodies
- 25. History substance and/or alcohol abuse or dependence within the past 1 year, at the investigator's judgment
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision)
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4 or 5 on the C-SSRS
- 31. Current or pending incarceration
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness

### 4.6 Concomitant Medications

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Patients should stay on stable regimen of other concomitant medications for the treatment of SLE (eg, analgesics, NSAIDs, statins, ACE inhibitors/ARBs and other antihypertensive drugs), unless changes in these treatments are

clinically indicated. Use of any other drugs for non-SLE conditions, including over-the-counter medications and herbal preparations, should remain stable unless change or addition is clinically necessary. Discussion with the medical monitor prior to initiation of new medication is strongly recommended. Any concomitant therapies must be recorded on the eCRF. Prior and concomitant medication use will be recorded for the 30 days prior to screening until the last follow-up visit. In addition, historical treatment for SLE (including immunosuppressant, anti-malarial, corticosteroid, and/or biologic agent) will be recorded for the 48 weeks prior to screening in the eCRF.

#### 4.6.1 Oral Corticosteroid Dose

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day).

After Day 0 (after initiation of study therapy), no up-titration above 10 mg/day is allowed except for up to 1 CS burst for increased disease activity.

Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits.

- Once a patient has received the first dose of study drug, prednisone (or prednisone equivalent) may be tapered down at the discretion of the investigator
  - Tapering is allowed after randomization except within 60 days of the primary (Day 210) and secondary (Day 120) endpoint assessments. Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant.

A maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed during the study between Day 0 and Day 60, according to the following:

- An oral CS "burst" between Day 0 and Day 60; (an increase of ≤ 40 mg/day of prednisone or equivalent), which must be tapered down to a maximum of 10 mg/day within 2 weeks of initiation of the "burst"
  - Alternatively, a single intramuscular (IM) dose of methylprednisolone (40 mg or equivalent) is permitted
  - o The course of the oral CS "burst" is not permitted to extend beyond Day 60

Treatment with inhalational CS therapy (eg, for asthma), or by any other route, is allowed. Other concomitant medications for SLE need to be taken at stable doses as per the inclusion criteria (Section 4.4).

### 4.6.2 Other Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in APPENDIX 4. Medications taken within 30 days prior to screening must be recorded on the eCRF.

- 1. Prior exposure to BOS161721
- 2. Patients who have received treatment with anti-CD20 monoclonal antibodies within 6 months of screening; recovery of B cells (CD19+) must be documented (record absolute number of CD19+ B cells)
- 3. Patients who have received treatment with cyclophosphamide within the 1 year prior to screening
- 4. Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria (oral or topical) within 3 months of screening
- 5. Patients who are currently receiving or are scheduled to receive plasmapheresis or lymphapheresis therapy, or have received such therapy within 8 weeks prior to screening
- 6. Patients who have received any live vaccines within 30 days of screening. Note: Furthermore, live vaccines should not be used during the course of the study and within the 2 months following last dose. Other inactivated vaccines such as tetanus, etc, may be used according to local guidelines during treatment period
- 7. Patients who are scheduled or anticipated to have elective surgery during the course of the study
- 8. Initiation of new immunosuppressant or anti-malarial agent is not permitted. Note: Dose reduction or replacement may be allowed due to intolerability or shortage for patients on a stable dose prior to study initiation

# 4.7 Women of Childbearing Potential

WOCBP is defined as any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) and is not postmenopausal.

See Section 4.7.2 for detailed information regarding contraceptive requirements for WOCBP.

# **4.7.1 Determination of Menopause**

Menopause is defined as at least 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes. Women under the age of 55 years must have a documented serum FSH level > 40 mIU/mL at screening to confirm menopause.

# 4.7.2 Contraception

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion.

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion.

Investigators shall counsel WOCBP and men who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and men who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, patients must agree to the use of 1 method of highly effective contraception from the following:

- Male condoms with spermicide
- Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as 1 of the acceptable methods of contraception since they will not be receiving study drug.
- IUDs, such as ParaGard®
- Vasectomy
- Complete abstinence, defined as complete avoidance of heterosexual intercourse, is an
  acceptable form of contraception. Women who are abstinent while participating in the study
  must continue to have pregnancy tests. Acceptable alternate methods of highly effective
  contraception must be discussed in the event that the patient chooses to forego complete
  abstinence.

Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing.

# 4.8 Deviation from Inclusion/Exclusion Criteria

Deviation from the inclusion or exclusion criteria will not be allowed. If deviation of inclusion/exclusion criteria is discovered after randomization, the investigator should contact the medical monitor for discussion. A decision will be made whether to allow a patient continue or withdrawal from the study medication.

See Section 6.8 for additional details.

# 4.8.1 Patient Withdrawal and Replacement

See Section 5.5 for reasons for removal from the trial. Withdrawn patients may be replaced during the MAD study after discussion between the principal investigator or designee and sponsor.

## 5 STUDY PROCEDURES

Refer to the eCRF completion guidelines for data collection requirements and documentation of study assessments/procedures.

# 5.1 Screening

Screening will be the same for both the MAD and POC studies.

Screening will take place from Day -28 to Day -1, and assessments may be performed over more than 1 visit. Confirmation that the most current IRB/IEC approved informed consent form (ICF) has been signed must occur before any study-specific screening procedures are performed. Procedures that are part of standard of care are not considered study-specific procedures and may be performed prior to informed consent and used to determine eligibility.

All screened patients will be assigned a unique screening number. The screening number will include a 3-digit site number and a 4-digit sequential number to identify patients from the time of screening. Only eligible patients who are confirmed by central review as meeting the inclusion/exclusion criteria, listed in Section 4.4 and Section 4.5 respectively, will be enrolled in the study. Screened patients who drop out of the clinical study before randomization will be recorded as screen failures. If rescreening occurs, the site will assign a new screening number.

Specific procedures at the screening visit will include:

- Medical history documentation
- Review of inclusion and exclusion criteria
  - o Patient medical records must contain documentation of SLE diagnosis
  - o C-SSRS
- Concomitant medication documentation
- Demographics
- Full physical examination
- Vital signs
- Chest x-ray
- Laboratory evaluations (nonfasting):
  - o Hematology and clinical chemistry
  - o Serology (Hepatitis B and C; HIV-1/2 combination)
  - o TB test
  - o CRP

- o Direct Coomb's test (if indicated for hemolytic anemia)
- o CD4+ count, total IgG and IgM levels, plasma CC , CCl
- Serum pregnancy test (WOCBP)
- o FSH (postmenopausal women)
- o Spot urine for protein/creatinine ratio
- o Urinalysis
- Stool sample
- 12-lead ECG
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, Physician's Global Assessment (PGA) of disease activity

Screening procedures are listed in the Schedule of Assessments (Section 3.4), and details are provided in Section 6.

### **5.1.1** Retesting During Screening Period

A single retesting of laboratory parameters and/or other assessments during the screening period is permitted (in addition to any parameters that require a confirmatory value) only if:

- medically indicated
- there is evidence a laboratory sample was mislabeled, indeterminate, inadequately processed, and/or deteriorated in transit to the central laboratory

Any new result will override the previous result (ie, the most current result prior to randomization) and is the value by which study inclusion/exclusion will be assessed, as it represents the patient's most current clinical state. This will also apply to patients who are being rescreened.

# 5.2 Enrollment/Randomization and Day 0 Treatment

Randomization should occur after patient eligibility for enrollment has been confirmed by the central eligibility review.

The study site will obtain a randomization number when registering the patient in IWRS. All patients will receive BOS161721 or placebo according to the kit number assigned by the IWRS randomization scheme.

After randomization, procedures include:

- PROs: CC
- C-SSRS
- Laboratory evaluations (fasting):
  - o Hematology and clinical chemistry
  - o Direct Coomb's test (if indicated for hemolytic anemia)


- CD4+ count, total IgG and IgM levels, plasma CCl , plasma CCl , whole blood for leukocyte immunophenotype
- o ADA
- o pSTAT3 (predose [trough] samples only in Phase 1b)
- o CCI
- o CCI
- o See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies
- o Urine pregnancy test will be collected on WOCBP prior to study drug administration
- o Spot urine for protein/creatinine ratio
- Urinalysis
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Full physical examination
- Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours postdose on Day 0)
- 12-lead ECG (prior to PK blood draw)
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, PGA)
- SLICC/ACR damage index
- Study drug administration:
  - Administration of BOS161721 or placebo will take place on-site, and is discussed in Section 7.3
- Injection site reaction assessment performed at 2 hours postdose

Procedures on Day 0 are listed in the Schedule of Assessments (Section 3.4), and details are provided in Section 6.

All patients who are enrolled, randomized, and receive study drug, or undergo study-specific procedures should reconsent with any updated versions of IRB/IEC approved informed consents during study participation as applicable and per institutional guidelines.

# 5.3 Treatment Period/Follow-Up Visits

The following procedures will be performed as indicated in the Schedule of Assessments (Table 1 and Table 2). See Schedule of Assessment tables for allowable windows for each visit.

- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- PROs: CC
- Urine pregnancy tests will be collected on WOCBP prior to study drug administration
- Injection site reaction assessments will be performed predose


- Direct Coomb's test (if indicated for hemolytic anemia)
- Spot urine for protein to creatinine ratio
- Urinalysis
- · CCI
- Plasma CCI
- PGA, BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, and the CLASI will be completed
- SLICC/ACR Damage Index will be completed at Day 180
- C-SSRS
- ECGs prior to PK blood draw
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies, respectively
- Fasting hematology and chemistry assessments
- The CD4+ count and total IgG and IgM levels
- Plasma **CC** & **CC**, ADA, and whole blood for leukocyte immunophenotype
- pSTAT3 (predose [trough] samples only Phase 1b)
- CRP and nAb will be assessed if patient is positive for ADA
- CCI

# 5.4 Safety Follow-Up Visits

Safety follow-up visits will take place at Days 210, 240, and 270. These visits will include the following assessments as indicated in the Schedule of Assessments (Table 1 and Table 2):

- PROs: CC
- Documentation of AEs and SAEs (see Section 6.2.2.5 on SAE reporting requirements)
- Injection site reactions
- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Spot urine for protein/creatinine ratio and urinalysis
- Concomitant medication documentation
- BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, and PGA
- Fasting clinical laboratory assessments (hematology and clinical chemistry)
- Direct Coomb's test (if indicated for hemolytic anemia)
- Plasma **CC**
- · CCI
- 12-lead ECG (prior to PK blood draw)
- CRP
- ADA
- CCI


• See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies, respectively

### 5.5 Premature Discontinuation

While patients are encouraged to complete all study evaluations, they may withdraw from the study at any time and for any reason. Every effort will be made to determine why any patient withdraws from the study prematurely. If the patient is unreachable by telephone, a registered letter, at the minimum, should be sent to the patient requesting him/her to contact the clinic.

All patients who withdraw from the study with an ongoing AE or SAE must be followed until the end of study or until the event is resolved or deemed stable, respectively.

If a patient withdraws prematurely after dosing, an end of treatment (EOT) visit should be performed (Day 180) and a last follow-up visit 90 days after dosing should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 5.4).

Patient participation may be terminated prior to completing the study and the reason recorded as follows:

- AE/SAE
- Protocol deviation
- Lost to follow-up
- Patient withdraws consent at their own request
- Investigator decision
- Decision by sponsor (other than AE/SAE, protocol deviation, or lost to follow-up)

Withdrawn patients may be replaced after discussion between the investigator or designee and sponsor.

# 6 ASSESSMENTS

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances, outside of the control of the investigator, which may make it unfeasible to perform the test. In these cases, the investigator will take all steps necessary to ensure the safety and wellbeing of the patient. When a protocol required test cannot be performed the investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. All protocol violations are entered directly into the eCRFs.

# 6.1 Medical History, Demographic and Other Baseline Information

The medical history comprises:

General medical history


- Documentation of SLE diagnosis
- Historical medication therapy for SLE

The following demographic information will be recorded:

- Age
- Ethnic origin (Hispanic/Latino or not Hispanic/not Latino)
- Race (White, American Indian/Alaska Native, Asian, Native Hawaiian or other Pacific Islander, Black/African American)
- Height (without shoes, in cm)
- Body weight, without shoes (kg)
- Body mass index (BMI [kg/m<sup>2</sup>])

Other baseline characteristics will be recorded as follows:

- Concomitant medication documentation (see Section 4.6)
- Status of child bearing potential and contraception

# **6.2** Safety Assessments

# **6.2.1** Laboratory Assessments

Laboratory tests will be performed at times defined in the Schedule of Assessments (Section 3.4). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

A central laboratory will be used (with the exception of urine pregnancy tests and stool analysis) to ensure accuracy and consistency in test results. The central laboratory will transmit all results for protocol tests, scheduled and unscheduled, to the clinical data base. Laboratory/analyte results that could unblind the study (ie, biomarker results) will not be reported to investigative sites. Urinalysis will be performed on midstream, clean catch specimens. Some biomarkers listed above will not be drawn at some sites due to geographical logistical challenges. See the laboratory manual for details.

Endpoint analyses will be based on changes from baseline assessments at Days 120 and 210.


**Table 3.** Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| Hemoglobin | BUN | рН | Spot urine for protein/creatinine ratio |
| Hematocrit | Creatinine | Glucose (qual) | FSH <sup>b</sup> |
| RBC count | Glucose (fasting) | Protein (qual) | Urine pregnancy test <sup>c</sup> |
| RDW | Calcium | Blood (qual) | QuantiFERON®-TB Gold In-Tube test |
| MCV | Sodium | Ketones | (QFT-G) |
| MCH | Potassium | Nitrites | Serology <sup>d</sup> (Hepatitis B and C; HIV-1/2 |
| MCHC | Chloride | Leukocyte esterase | combination) |
| Platelet count | Total CO <sub>2</sub> (bicarbonate) | Urobilinogen | Stool sample <sup>e</sup> |
| WBC count | AST, ALT | Urine bilirubin | |
| CD4+ count | Total bilirubin | Microscopy <sup>a</sup> | |
| Total neutrophils | Alkaline phosphatase | | |
| (Abs) | Creatine kinase | | |
| Eosinophils (Abs) | Uric acid | | |
| Monocytes (Abs) | Albumin | | |
| Basophils (Abs) | Total cholesterol | | |
| Lymphocytes (Abs) | (fasting) | | |
| | LDL-C (fasting) | | |
| | HDL-C (fasting) | | |
| | Triglycerides (fasting) | | |
| | Total protein | | |
| | PT/INR | | |
| | Additional Tests <sup>f</sup> | | Immunogenicity, PD and other |
| | (potential Hy's Law) | | Biomarker Tests |
| | AST, ALT (repeat) | | ADA |

| Additional Tests <sup>1</sup> | Immunogenicity, PD and other |
|-------------------------------|----------------------------------|
| (potential Hy's Law) | Biomarker Tests |
| AST, ALT (repeat) | ADA |
| Total bilirubin (repeat) | $nAb^g$ |
| Albumin (repeat) | pSTAT3 (predose [trough] samples |
| Alkaline phosphatase | only in Phase 1b) |
| (repeat) | Total IgG & IgM |
| Direct bilirubin | Plasma CCI |
| Indirect bilirubin | Plasma CCI & CCI |
| GGT | Whole blood for leukocyte |
| | immunophenotype |
| | CCI |
| | CCI |
| | CCI<br>CCI<br>CCI |
| | CRP |
| | Direct Coomb's test <sup>h</sup> |

Abbreviations: Abs = absolute; ADA = anti-drug antibody; ALT = alanine aminotransferase;

; CCl ; AST = aspartate aminotransferase; BUN = blood urea

nitrogen; C = complement; CD4+ = cluster of differentiation 4; CRP = C-reactive protein;

dsDNA = double-stranded deoxyribonucleic acid;; FSH = follicle stimulating hormone;

GGT = gamma-glutamyltransferase; HDL-C = high-density lipoprotein cholesterol; HIV = human

immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; INR = international normalized

ration; IL-21 = interleukin 21; LDL-C = low-density lipoprotein cholesterol; MCH = mean corpuscular

hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = Mean corpuscular volume;

nAb = neutralizing antibody; pSTAT3 = phosphorylated signal transducer and activator of transcription 3;

PT = prothrombin time; qual = qualitative; RBC = red blood cell; RDW = RBC distribution width; SAE = serious


Table 3. Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests | Other Safety Tests |
|---|---|---|---|---|
| adverse event; SC = | subcutaneous; CCI | | ; | TB = tuberculosis. |

- a. On all urine samples.
- b. At screening only, in women who are amenorrheic for at least 12 consecutive months and under 55 years old.
- c. For WOCBP.
- d. Screening only.
- e. At screening, and if a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- f. Additional testing for potential Hy's Law cases only (See Section 6.2.2.6.3).
- g. If patient is positive for ADA.
- h. If clinically indicated for hemolytic anemia.

# 6.2.1.1 Pregnancy testing

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 5.4).

See Section 6.2.2.7.1 for information on reporting of pregnancies as AEs/SAEs during the study.

## **6.2.1.2** Tuberculosis Screening

During the screening period, it must be determined and documented that a patient does not have evidence of active or latent or inadequately treated TB per the exclusion criteria (Section 4.5). The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).

# 6.2.1.2.1 Mycobacterium Tuberculosis Testing Using QuantiFERON Test<sup>40</sup>

QuantiFERON®-TB Gold In-Tube (QFT-G) is an in vitro diagnostic test using a peptide cocktail simulating ESAT-6, CFP-10, and TB 7.7 proteins to stimulate cells in heparinized whole blood. Detection of INFγ performed by enzyme-linked immunosorbent assay (ELISA) is used to identify in vitro responses to these peptide antigens that are associated with Mycobacterium tuberculosis infection. QFT-G is an indirect test for M. tuberculosis infection (including disease) and is intended for use in conjunction with risk assessment, radiography and other medical and diagnostic evaluations.

Test results will be reported as positive, negative, or indeterminate. A negative QFT-G test result is required to meet the inclusion criterion. In the case of an indeterminate result, repeat tests should be permitted for the purpose of determining eligibility of patients to enroll in this study. If a repeat test is indeterminate again, the patient is a screen failure. The procedure for using this test and interpreting the results will be described fully in the laboratory manual, which will be provided to investigators.

#### **6.2.2** Adverse Events

#### 6.2.2.1 Definitions

An AE is defined as any untoward medical occurrence experienced by a study patient, whether or not considered drug related by the principal investigator.

AEs are unfavorable changes in a general condition, subjective or objective signs or symptoms, worsening of pre-existing concomitant disease, and clinically significant abnormality in laboratory parameters observed in a patient in the course of a clinical study.

Non-serious SLE manifestations or abnormal laboratory results related to SLE disease activity would not be recorded as AEs unless they meet the definition for SAEs (Section 6.2.2.5).

## **6.2.2.2** Recording of Adverse Events

AEs should be collected and recorded for each patient from the date of the first dose of study drug until the end of their participation in the study, including the safety follow up period.

AEs may be volunteered spontaneously by the study patient, or discovered by the study staff during physical examinations or by asking an open, nonleading question such as 'How have you been feeling since you were last asked?' All AEs and any required remedial action will be recorded on the Adverse Events eCRF and Safety Adverse Event Form. The details of the AE, date of AE onset (and time, if known), date of AE outcome (and time, if known), and action taken for the AE will be documented together with the principal investigator's assessment of the seriousness of the AE and causal relationship to the study drug and/or the study procedure.

All AEs should be recorded individually, using diagnostic terms where possible. If the diagnosis is not established, individual symptoms may be reported. The AEs will subsequently be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

### **6.2.2.3** Severity of Adverse Events

Each AE will be assessed by the principal investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 criteria. <sup>41</sup> When changes in the severity (grade) of an AE occur more frequently than once a day, the maximum severity for the event should be noted for that day. Any change in severity of signs and symptoms over a number of days will be captured by recording a new AE, with the amended severity grade and the date (and time, if known) of the change.


# **6.2.2.4** Causality of Adverse Events

The principal investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (Table 4) should be selected based on medical judgment, considering the definitions below and all contributing factors.

| Table 4. | Causality Definitions |
|---|---|
| Related | A clinical event, including laboratory test abnormality, occurs in a plausible time relationship to treatment administration and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (dechallenge <sup>a</sup> ) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge <sup>b</sup> procedure if necessary. |
| Unrelated | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative dechallenge and rechallenge information. Typically explained by extraneous factors (eg, concomitant disease, environmental factors, or other drugs or chemicals). |

Dechallenge: Upon discontinuation of a drug suspected of causing an AE, the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation (positive dechallenge), or the symptoms continue despite withdrawal of the drug (negative dechallenge). Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia).

An unexpected adverse drug event is any adverse drug event for which the specificity or severity is not consistent with the current IP.

### **6.2.2.5** Seriousness of Adverse Events

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life threatening; this means that the patient was at risk of death at the time of the event; it does not mean that the event hypothetically might have caused death if it were more severe
- Requires hospitalization or prolongation in existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly or birth defect
- Is another important medical event (see below)

Important medical events that do not result in death, are not life threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such events are:

Rechallenge: Upon re-administration of a drug suspected of causing an AE in a specific patient in the past, the AE recurs upon exposure (positive rechallenge), or the AE does not recur (negative rechallenge).
BOS161721


- Intensive treatment in an emergency room or at home for allergic bronchospasm
- Blood dyscrasias or convulsions that do not result in inpatient hospitalization
- Development of drug dependency or drug abuse

Hospitalization for elective surgery or routine clinical procedures that are not the result of AE (eg, elective surgery for a pre-existing condition that has not worsened) need not be considered SAEs. If anything untoward is reported during the procedure, that occurrence must be reported as an AE, either 'serious' or 'nonserious' according to the usual criteria.

Suspected unexpected serious adverse reactions (SUSARs) are AEs that are associated with the use of the drug and are serious and unexpected.

# **6.2.2.6** Adverse Events of Special Interest

AEs of special interest in this study include the following:

- 1. Anaphylaxis and serious allergic reactions
- 2. Grades 2 to 5 injection site reaction, including erythema, pain, and induration (See APPENDIX 6)
- 3. Drug Induced Liver Injury (DILI) assessed following Hy's Law
- 4. Malignancy
- 5. Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, and disseminated tuberculosis
- 6. Cryptosporidiasis

# 6.2.2.6.1 Anaphylaxis and Serious Allergic Reactions

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria. <sup>42</sup> In the event of anaphylactic reaction or severe/serious hypersensitivity/allergic reaction, the patient must discontinue IP and emergency resuscitation measures implemented. In case of other mild to moderate hypersensitivity reaction, depending on the severity, the investigator may manage in accordance with the standard-of-care.

Anaphylaxis is highly likely when any one of the following 3 criteria is fulfilled:

- 1. Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (eg, generalized hives, pruritus, or flushing, swollen lips-tongue-uvula) and at least 1 of the following:
  - a. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow [PEF], hypoxemia)
  - b. Reduced blood pressure or associated symptoms of end-organ dysfunction (eg, hypotonia [collapse], syncope, incontinence)

- 2. Two or more of the following that occur rapidly after exposure to a likely allergen for that patient (minutes to several hours):
  - a. Involvement of the skin-mucosal tissue (eg, generalized hives, itch-flush, swollen lips-tongue-uvula)
  - b. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)
  - c. Reduced blood pressure or associated symptoms (eg, hypotonia [collapse], syncope, incontinence)
  - d. Persistent gastrointestinal symptoms (eg, crampy abdominal pain, vomiting)
- 3. Reduced blood pressure after exposure to known allergen for that patient (minutes to several hours):
  - a. Systolic blood pressure of less than 90 mm Hg or greater than 30% decrease from the patient's baseline

# 6.2.2.6.2 Injection Site Reactions

Injection site reactions are to be captured and reported as AEs. These will include Grades 2 to 5 injection site erythema, pain, and induration (see APPENDIX 6). The investigator should provide a clear description of the observed or reported AE including location and severity. All concomitant treatments used to treat injection site reactions should be recorded and captured in the eCRF, together with the AE of injection site reactions.

# 6.2.2.6.3 Potential Drug-Induced Liver Injury

Abnormal values in AST and/or ALT levels concurrent with abnormal elevations in total bilirubin level that meet the criteria outlined below in the absence of other causes of liver injury are considered potential cases of DILI, and as potential Hy's Law cases, and should always be considered important medical events. If symptoms compatible with DILI precede knowledge of serum chemical test abnormalities, liver enzyme measurements should be made immediately, regardless of when the next visit or monitoring interval is scheduled. In some cases, symptoms may be an early sign of injury and although typically less sensitive than serum enzyme elevations, they may indicate a need for prompt serum testing. An increase in liver enzymes should be confirmed by a repeated test within 48 to 72 hours following the initial test, prior to reporting of a potential DILI event. Patients will continue to have weekly or biweekly liver enzyme measurements until resolution or levels return to baseline.

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 6.2.2.7.2 for reporting details).

Potential DILI is defined as:

1. ALT or AST elevation  $> 3 \times ULN$ 

**AND** 

2. Total bilirubin > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)

#### AND

3. No other immediately apparent possible causes of ALT or AST elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic

The patient should return to the investigational site and be evaluated as soon as possible, include laboratory tests, detailed history, and physical assessment. In addition to repeating measurements of AST and ALT, laboratory tests should include albumin, CK, total bilirubin, direct and indirect bilirubin, GGT, prothrombin time (PT)/International Normalized Ratio (INR), and alkaline phosphatase. A detailed history, including relevant information, such as review of ethanol, acetaminophen, recreational drug and supplement consumption, family history, occupational exposure, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and work exposure, should be collected. Further testing for acute hepatitis A, B, or C infection and liver imaging (eg, biliary tract) may be warranted. All cases confirmed on repeat testing as meeting the laboratory criteria defined above, with no other cause for liver function test (LFT) abnormalities identified at the time should be considered potential Hy's Law cases irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal LFTs. Such potential Hy's Law cases should be reported as SAEs.

Study drug discontinuation is considered if there is marked serum AST or ALT elevation or evidence of functional impairment (as indicated by rising bilirubin or INR, which represent substantial liver injury) that is related to study drug. Discontinuation of treatment should be considered if:

- ALT or AST > 8 × ULN
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks

Discontinuation of treatment must occur if:

- ALT or AST >3 × ULN and (total bilirubin > 2 × ULN or INR > 1.5)
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%)

# *6.2.2.6.4 Malignancy*

The identification of a malignancy event will be made by the study site and communicated to the sponsor or designee. AEs should be reported as serious per the criteria in Section 6.2.2.5.

After the first dose of study drug, when there is a decision to biopsy a potentially malignant tumor, lymph node, or other tissue, the investigator and/or consultant(s) should contact the sponsor clinicians or designee to discuss the issue and any decisions as soon as possible.

# 6.2.2.6.5 Specific Infections

Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, shingles, disseminated herpes simplex, or disseminated tuberculosis will be recorded as AEs of special interest.

Cryptosporidiosis is also considered an AE of special interest. Patients will be evaluated for cryptosporidium in the stool at screening, and as clinically indicated (eg, watery diarrhea) during the study. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

# **6.2.2.7** Reporting of Adverse Events

AE reporting will be carried out in accordance with applicable local regulations, including regulatory agency and IRB reporting requirements.

Each AE is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

# 6.2.2.7.1 Reporting of Pregnancy

As information is available, a pregnancy diagnosed during the study will be reported within 24 hours to the sponsor via the Pregnancy Notification and Outcome Form, including pregnancy in female patients who received study drug and female partners of male study patients who received study drug. The pregnancy should be followed to term and/or outcome and this outcome should also be reported to the sponsor via the Pregnancy Notification and Outcome Form. Pregnancy itself is not regarded as an AE or SAE unless there is complication.

In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an AE or SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live born, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as serious adverse events when the investigator assesses the neonatal death as related or possibly related to exposure to investigational product.

# 6.2.2.7.2 Reporting of Serious Adverse Events

The principal investigator is responsible for providing notification to the sponsor of any SAE via the Safety Adverse Event Form, whether deemed study drug related or not, that a patient experiences during their participation in this study within 24 hours of becoming aware of the event.

If an SAE is fatal or life threatening, notification to the sponsor must be made aware immediately, irrespective of the extent of available AE information. This timeframe also applies to additional new information (follow-up) on previously forwarded SAE reports as well as to the initial and follow-up reporting of exposure during pregnancy and exposure via breastfeeding cases. In the rare event that the investigator does not become aware of the occurrence of an SAE immediately (eg, if an outpatient study patient initially seeks treatment elsewhere), the investigator is to report the event within 24 hours after learning of it and document the time of his/her first awareness of the AE.

The principal investigator will review each SAE and evaluate the intensity and the causal relationship of the event to the study drug. All SAEs will be recorded from the time of first dose of study drug through the safety follow-up period (up to Day 270). SAEs occurring after the final follow-up visit and coming to the attention of the principal investigator must be reported only if there is (in the opinion of the principal investigator) reasonable causal relationship with the study drug.

As a minimum requirement, the initial notification should provide the following information:

- Study number
- Patient number
- Details of the SAE (verbatim details are sufficient for immediate notification)
- Criterion for classification as 'serious'
- Causality assessment (which may be updated in a follow-up report when sufficient information is available to make this classification)

Initial reports of SAEs must be followed later with detailed descriptions, including clear photocopies of other documents as necessary (eg, hospital reports, consultant reports, autopsy reports, etc), with the study patient's personal identifiers removed. All relevant information obtained by the principal investigator through review of these documents will be recorded and submitted to the sponsor within 24 hours of receipt of the information. If a new Safety Adverse Event Form is submitted, then the principal investigator must sign and date the form. The sponsor may also request additional information on the SAE, or clarification of omitted or discrepant information from the initial notification, which the principal investigator or an authorized delegate should submit to the sponsor within 24 hours of the request as possible.

# 6.2.2.7.3 Reporting of Adverse Events of Special Interest

AEs of special interest will be reported to safety immediately or within 24 hours of the site becomes aware of the event and recorded as such on the Adverse Events eCRF and Safety Adverse Event Form.

Potential DILI will be reported based on specifications mentioned in Section 6.2.2.6.3.

Each AE of special interest is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 6.2.2.7.2.

#### **6.2.2.8** Follow Up of Adverse Events

All AEs will be followed up through the safety follow-up visits. All SAEs experienced by a patient, irrespective of the suspected causality, will be monitored until the event has resolved, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the principal investigator and medical monitor, until there is a satisfactory explanation for the changes observed, or until the patient is lost to follow-up.

See Section 6.2.2.7.1 for details related to follow-up of pregnancy. See Section 6.2.2.6.3 for details related to follow-up of potential DILI. See Section 6.2.2.6.4 for details related to follow-up of malignancy.

#### 6.2.3 Vital Signs

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (Section 3.4). Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq 5$  minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

# 6.2.4 12-Lead Electrocardiograms

ECG will be assessed as specified in the Schedule of Assessments (Section 3.4). ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

The ECG will include all 12 standard leads and a Lead II rhythm strip on the bottom of the tracing. The ECG will be recorded at a paper speed of 25 mm/second. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QT interval corrected for heart rate using Fridericia's formula (QTcF).

All ECGs must be evaluated by a qualified physician or qualified designee for the presence of abnormalities and will be captured electronically and retained for future evaluation if required, up to the time of the clinical study report (CSR) completion.

#### 6.2.5 Physical Examinations

The full physical examination will be completed at screening and Day 0. It includes an assessment of general appearance and evaluation of head, eyes, ears, nose, mouth, throat, neck,

thyroid, lymph nodes, and extremities, and dermatologic, respiratory, cardiovascular, gastrointestinal, musculoskeletal, neurologic, and psychiatric systems.

The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Section 3.4). It includes evaluation of patient complaints and SLE disease-related issues, and will exclude the genitourinary system.

#### 6.2.6 C-SSRS

The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed by Columbia University researchers for the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening.<sup>43</sup>

The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Section 3.4). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

# **6.2.7** Injection Site Reactions

Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (Section 3.4). Local injection site reactions will be assessed at 2 hours postdose at baseline, and predose for each injection after baseline. Injection site reactions should be managed according to the standard of care. Injection site reactions, Grades 2 to 5, are to be reported as AEs of special interest (see Section 6.2.2.7.3).

#### 6.2.8 Immunogenicity

The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (Section 3.4). Blood samples (4 mL) to provide approximately 1.5 mL of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K<sub>2</sub>EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.

After the first dose, if a patient tests positive in the validated confirmatory ADA assay, the sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay.

# **6.3** Efficacy Assessments

All efficacy assessments will be performed at times defined in the Schedule of Assessments (Section 3.4).

#### **6.3.1 SLEDAI-2K**

The SLEDAI-2K is a validated instrument that measures disease activity in SLE patients at the time of the visit and in the previous 30 days. It is a global index and includes 24 clinical and laboratory variables that are weighted by the type of manifestation, but not by severity. The total score falls between 0 and 105, with higher scores representing increased disease activity. The SLEDAI-2K has been shown to be a valid and reliable disease activity measure in multiple patient groups. A SLEDAI -2K of 6 or more generally represents moderately to severely active disease. 44

#### 6.3.2 BILAG 2004

The BILAG-2004 index is an organ-specific 97-question assessment based on the principle of the doctor's intent to treat. Only clinical features attributable to SLE disease activity are to be recorded and based on the patient's condition in the last 4 weeks compared with the previous 4 weeks. It will be scored as not present (0), improved (1), the same (2), worse (3), or new (4). Disease activity is graded separately for 9 body systems to 5 different grades (A to E) as follows: A ("Active") is very active disease, B ("Beware") is moderate activity, C ("Contentment") is mild stable disease, D ("Discount") is inactive now but previously active, and E ("Excluded") indicates the organ was never involved. A shift from BILAG-2004 Grade A or B to a lower grade indicates a clinically relevant change in disease activity as the BILAG-2004 grades mirror the decision points for treatment interventions.

Only investigators that complete BILAG-2004 training will be allowed to perform the BILAG-2004 assessments. Preferably, the same investigator should evaluate the patient at each BILAG-2004 assessment from screening to study completion. The investigator must maintain documentation with descriptive details supporting the BILAG-2004 scoring (eg, chart, worksheet, clinic notes, and labs) at each visit.

See APPENDIX 5 for detailed specifications.

#### 6.3.3 PGA of Disease Activity

The PGA is used to assess investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients".

When scoring the PGA, the assessor should always look back at the score from the previous visit.

# 6.3.4 Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response

# **6.3.4.1 SRI-4 Response**

The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. Response based on the SRI-4 is defined by:

1)  $\geq$  4-point reduction in SLEDAI-2K global score, 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B), and 3) no deterioration from baseline in the PGA by  $\geq$  0.3 points. The SRI-4 response in patients with moderate to severe SLE is associated with broad improvements in clinical and patient-reported outcomes. <sup>45</sup>

# 6.3.4.2 SRI-5 and SRI-6 Response

Like the SRI-4, the SRI-5 and SRI-6 are composite indices of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. However, the SRI-5 and SRI-6 are computed with a minimal three-point or five-point improvement in SLEDAI-2K being required, respectively.<sup>46</sup>

# 6.3.4.3 BICLA Response

The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and PGA. BICLA response is defined as 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (eg, all B [moderate disease] scores falling to C [mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4)  $\leq$  10% deterioration in PGA score and 5) no treatment failure. 44 It is driven primarily by the BILAG, and has been used in Phase 2 and 3 mAb studies. 47

For the endpoints of BICLA response at Days 210, 240, and 270, patient scores will be completed and response determined.

#### 6.3.5 CLASI Response

The CLASI is a comprehensive tool for assessment of disease activity and damage in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity. <sup>48</sup> Response is defined as 50% improvement from baseline in "A" or "B" scores. This assessment will be applied to all patients as all are required to have cutaneous disease activity.

For the secondary efficacy endpoint of CLASI response at Day 210, patient scores on MAD and POC studies will be compared with baseline for 50% improvement.

#### 6.3.6 ACR-28 Joint Count

The ACR-28 joint count will evaluate the number of tender and swollen joints in the shoulder, elbow, wrist, hand, knee joints. Joints of the feet are excluded.

#### 6.4 Other Variables

#### 6.4.1 SLICC/ACR Damage Index

The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in patients with SLE regardless of cause, with demonstrated content, face, criterion, and discriminant validity. It will be performed on Days 0 and 180.

#### 6.4.2 **PROs**

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the CCI and the CCI and will be assessed as specified in the Schedule of Assessments (Section 3.4).



#### 6.5 Pharmacokinetic Assessments

During the MAD Phase 1b (all sites) and POC Phase 2 (select sites only) studies, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to Table 1 and Table 2.

Plasma concentrations of BOS161721 will be measured using a validated immunoassay. The PK parameters will be calculated from the plasma concentration actual time profiles.

# 6.6 Pharmacodynamic Assessments

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (Section 3.4) for each of the following parameters:

- pSTAT3 (predose [trough] samples only Phase 1b)
- Antibodies: CCl
- Plasma complement (CCL)
- Plasma CCI and CCI
- Whole blood for leukocyte immunophenotype

# 6.7 Pharmacokinetic/Pharmacodynamic Relationship

Evidence of any PK/PD relationships will be evaluated between BOS161721 plasma concentrations and the available PD endpoints and biomarkers.

#### **6.8** Protocol Deviations

Protocol deviations will be documented during the study.

#### 7 STUDY DRUG MANAGEMENT

# 7.1 Description

#### 7.1.1 Formulation



Additional information regarding dose preparation will be provided in a separate Pharmacy Manual.

# **7.1.2 Storage**

All supplies of BOS161721 or placebo must be stored in accordance with the manufacturer's instructions. BOS161721 or placebo will be stored in a securely locked area, accessible to authorized persons only, until needed for dosing.

Information regarding storage and dose preparation will be provided in a separate Pharmacy Manual.

# 7.2 Packaging and Shipment

Investigational medicinal products will be supplied by Boston Pharmaceuticals, Inc. Investigational medicinal products will be packaged and labeled according to applicable local and regulatory requirements.

#### 7.3 Dose and Administration

Details of dosing are provided in Section 3.1.

Each unit dose will be prepared by a qualified staff member. The vials of investigational product (IP) will appear identical and will have a "blinded" label on the vials that will state mg or placebo. When the site goes into the IWRS to request the patient kit(s), the IWRS will assign the

BOS161721

appropriate number of kits (regardless of assignment to placebo or active treatment) per the dose (ie, CCI). If a patient is randomized to the placebo arm, they will receive the matching number of kits.

The designated staff member (or designee under the direction of the designated staff member) will dispense BOS161721 or placebo for each patient according to the protocol, randomization list, and Pharmacy Manual, if applicable.

After receiving sponsor approval in writing, the investigational site is responsible for returning all unused or partially used BOS161721 or placebo to the sponsor or designated third party or for preparing BOS161721 or placebo for destruction via incineration.

Further details are found in a separate Pharmacy Manual.

# 7.4 Accountability

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Products returned to the pharmacy will be stored under the same conditions as products not yet dispensed. The returned products should be marked as 'returned' and kept separate from the products not yet dispensed.

All dispensing and accountability records will be available for sponsor review after database lock procedures are completed. During safety monitoring, the drug accountability log will be reconciled with the products stored in the pharmacy.

# 7.5 Prohibited Concomitant Therapy

Prohibited concomitant medications are discussed in Section 4.6 and APPENDIX 4 and will be listed as protocol violations if taken when not permitted.

# 7.6 Compliance

Dosing will be performed by trained, qualified personnel designated by the principal investigator. The date and time of dosing will be documented on each dosing day. Comments will be recorded if there are any deviations from the planned dosing procedures.

#### **8 STATISTICS**

The following analyses are planned:

- An IA will be performed during the last cohort of the MAD phase to determine dose selection for the POC phase.
- The final analysis will be performed when all patients have completed the safety follow-up or withdrawn from the study.
- Safety analyses will be performed for DMC reviews throughout the study to evaluate dose escalation decisions and accumulating safety data. The frequency and details of the

content and format of the safety review meetings will be described in the SAP and/or DMC charter.

All statistical analyses will be performed using Statistical Analysis Software (SAS®) Version 9 or higher.

The following standards will be applied for the analysis unless otherwise specified. Data will be summarized descriptively by treatment and overall for each study phase. For the MAD phase, BOS161721 will be summarized overall and by each dose level, and placebo patients from each cohort will be combined. Select parameters will be summarized using patients from both study phases. Statistical testing will be performed on data from the Phase 2 study only.

Continuous data will be summarized using number, mean, standard deviation (SD), 25th and 75th percentiles, minimum, median, and maximum. Categorical data will be summarized by treatment group using frequency tables (number and percentage). Time to event data will be summarized using counts, medians, 25th and 75th percentiles, and standard error. All data will be listed for all patients.

Statistical inference will be based on a 2-tailed test with an overall 0.10 level of significance, unless stated otherwise.

The effects of noncompliance, background therapy use, treatment discontinuations, premature withdrawal from study and covariates will be assessed to determine the impact on the general applicability of results from this study. Exploratory analyses of the data will be conducted as deemed appropriate. Any deviations from the planned analyses will be described and justified in the final integrated CSR.

Protocol deviations and prohibited medications that define medication failures will be fully assigned and documented before database lock and unblinding.

Further details of the analysis, including the handling of missing data, transformations and other data handling procedures will be provided in the SAP.

# 8.1 Sample Size

Sample size in the Phase 1b study is based on operational consideration.

The sample size in the Phase 2 study is based on the primary endpoint, SRI-4 Response at Day 210. Approximately 156 additional patients will be randomized in a 2:1 ratio to BOS161721 versus placebo to achieve 132 evaluable subjects in the FAS. This assumes 24 subjects will drop prior to having received treatment and an evaluable post-baseline efficacy measure. Enrollment and randomization will be monitored in a blinded fashion and increased if needed to ensure at least 132 subjects are randomized into the FAS.

A total of 132 subjects randomized provides more than 80% power to detect a treatment difference of 25% in SRI-4 response rates at Day 210, based on a targeted 2-sided significance level of 10% and using a 2-sided Pearson's chi-squared test. This assumes of a response rate of 65% for BOS161721 and 40% for placebo, where missing data at Day 210 is carried forward

from most recent non-missing result and subjects are treated as a non-responder if a prohibited medication defined as a medication failure occurs.

#### **8.2** Statistical Methods

#### 8.2.1 Analysis Populations

The primary efficacy analysis will be based on the FAS, defined as all patients who receive at least 1 dose of study treatment and at have least 1 evaluable post-baseline efficacy evaluation. FAS analyses will be conducted on the basis of the randomized treatment.

A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be identified based on blinded data prior to study unblinding. PP analyses will be conducted on the basis of the randomized treatment.

Safety analyses will be based on the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. Safety analyses will be conducted on the basis of actual treatment received.

Pharmacokinetic analysis will be conducted on the PK analysis set, defined as the FAS with sufficient concentration data for the calculation of PK parameters.

#### 8.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized using all randomized patients.

#### 8.2.3 Primary Efficacy Endpoint(s)

The proportion of patients who achieve a SRI-4 response at Day 210 will be assessed via Pearson's chi-squared analysis. The primary efficacy endpoint will be analyzed using the FAS and if needed repeated in the PP analysis set. Missing values will be addressed by employing a last observation carried forward (LOCF) analysis. Other imputation methods may be employed as a sensitivity analysis and will be described in the SAP. Additional analyses exploring impact of baseline factors such as baseline disease severity, race, and other characteristics may be performed.

Patients that received prohibited medications or unallowable CS usage as described in Section 4.6 will be considered "medication failures" and will be treated as non-responders for the primary efficacy analysis. Patients that received an allowable CS burst but having missing data at Day 210 will considered a medication failure and will be treated as non-responders for the primary efficacy analysis. The determination of medication failures will be reviewed using blinded data and finalized prior to unblinding.

The superiority of BOS161721 relative to placebo will be evaluated. If the proportion of SRI-4 responders for the selected POC dose in BOS161721 arm is higher than that of the placebo arm, then BOS161721 will be considered superior to placebo if the 2-sided p-value is less than or

equal to 0.10. Secondary and exploratory endpoints for this POC study will be evaluated based on the same statistical hypothesis.

# 8.2.4 Secondary Efficacy Endpoint(s)

Binary efficacy endpoints will be assessed via Pearson's chi-squared analysis. Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) and treatment will be compared using the F-test. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test. The secondary efficacy endpoints will be analyzed on the FAS and if needed repeated in the PP analysis set. Details including handling of missing data and "medication failures" will be available in the SAP.

# 8.2.5 Analysis of Safety

# 8.2.5.1 Safety Analysis

Safety analyses will be performed on the SS. AE data will be coded to system organ class and preferred term using MedDRA. The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class an preferred term, will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be coded using the WHO Drug dictionary. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters will be summarized at each individual visit.

#### 8.2.6 Pharmacokinetic and Pharmacodynamic Data

# 8.2.6.1 Analysis of Pharmacokinetic Data

PK parameters will be calculated from concentration data collected during the MAD Phase 1b using non-compartmental analysis and include the following:

•  $C_{max}$ ,  $T_{max}$ , AUC,  $t_{1/2}$ , CL,  $V_{d}$ 

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:

- A listing of all plasma BOS161721 concentrations by patient at actual times post dose;
- A descriptive summary of plasma BOS161721 concentrations. Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.

#### 8.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Exploratory analyses examining the relationship between PD parameters and PK concentration and PK parameters will be performed.

# 8.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints.

# 8.3 Interim Analysis and Power

One IA is planned for this study and will be conducted at the time of the POC decision for dose selection.

Since there is no IA during the POC phase, there is no impact on the type 1 error.

#### 9 ETHICS AND RESPONSIBILITIES

#### 9.1 Good Clinical Practice

The procedures set out in this protocol are designed to ensure that the sponsor and the principal investigator abide by the principles of the International Council for Harmonisation (ICH) guidelines on GCP and the Declaration of Helsinki (Version 2013). The clinical study also will be carried out in the keeping with national and local legal requirements (in accordance with US IND regulations [21 CFR 56]).

#### 9.2 **DMC**

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for BOS161721. The recommendations made by the DMC (ie, dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.

The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the

accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) suggest dose for POC portion of the study as described in Section 3.1.1.3.

The DMC considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

The DMC will have access to unblinded treatment information during the clinical trial. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of BOS161721 treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.

# 9.3 Institutional Review Board/Independent Ethics Committee

Independent Ethics Committees (IEC)/Institutional Review Boards (IRB) must meet the guidelines set out by the U.S. Food and Drug Administration (FDA) and conform to local laws and customs where appropriate. Written IRB/IEC approval for the protocol and the signed ICF must be obtained and transmitted to Boston Pharmaceuticals or representative before the study can be initiated. The IRB/IEC must be informed of and approve all protocol amendments. The investigator will ensure that this study is conducted in full conformance with all applicable local and regional laws and regulations. The complete text of the World Medical Association Declaration of Helsinki is given in APPENDIX 2.

#### 9.4 Informed Consent

Before each patient undergoes any protocol required assessments or procedure, the written informed consent will be obtained according to the regulatory and legal requirements of the participating country. As part of this procedure, the principal investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study patient should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The principal investigator or designee will provide the sponsor with a copy of the IRB-approved ICF prior to the start of the study.

The informed consent document must be signed and dated; 1 copy will be handed to the patient and the principal investigator will retain a copy as part of the clinical study records. The principal investigator will not undertake any investigation specifically required for the clinical study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented.

If the informed consent document is revised, it must be reviewed and approved by the responsible IRB/IEC. Patients currently enrolled may need to sign this revision (based on IRB/IEC requirements) and all future patients enrolled in the clinical study will be required to sign this revised ICF.

# 9.5 Records Management

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes. The principal investigator or designee will cooperate with the sponsor's representative(s) for the periodic review of study documents to ensure the accuracy and completeness of the data capture system at each scheduled monitoring visit.

Electronic consistency checks and manual review will be used to identify any errors or inconsistencies in the data. This information will be provided to the respective study sites by means of electronic or manual queries.

The principal investigator or designee will prepare and maintain adequate and accurate study documents (medical records, ECGs, AE and concomitant medication reporting, raw data collection forms, etc.) designed to record all observations and other pertinent data for each patient receiving BOS161721 or placebo.

The principal investigator will allow sponsor representatives, contract designees, authorized regulatory authority inspectors, and the IRB to have direct access to all documents pertaining to the study.

Electronic case report forms are required and should be completed for each randomized patient. It is the principal investigator's responsibility to ensure the accuracy, completeness, legibility, and timeliness of the data reported on the patients' eCRF. Electronic case report forms should be completed in a timely fashion to support the study timelines. Source documentation supporting the eCRF data should indicate the patient's participation in the study and should document the dates and details of study procedures, AEs, and patient status. The principal investigator or designated representative should complete and the principal investigator should verify the source documents as the information is collected. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the Sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes.

#### 9.6 Source Documentation

The documents that will form the source data for the clinical study (eg, patient charts, laboratory reports) must be defined and documented in the in-house study master file prior to the start of the study. Data on the eCRFs which will be checked against source data during monitoring visits

must also be defined and documented in the in-house study master file including the percentage of each of the source data to be verified and the percentage of patients' eCRFs to be monitored.

#### 9.7 Study Files and Record Retention

According to ICH guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of BOS161721. However, these documents should be retained for a longer period if required by the applicable legal requirements.

#### 10 AUDITING AND MONITORING

Throughout the course of the study, the study monitor will make frequent contacts with the investigator. This will include telephone calls and on-site visits. The study will be routinely monitored to ensure compliance with the study protocol and the overall quality of data collected. During the on-site visits, the eCRFs will be reviewed for completeness and adherence to the protocol. As part of the data audit, source documents will be made available for review by the study monitor. The study monitor may periodically request review of the investigator study file to assure the completeness of documentation in all respects of clinical study conduct. The study monitor will verify that each patient has proper consent documentation from the patient and/or patient's authorized representative for study procedures and for the release of medical records to the sponsor, FDA, other regulatory authorities, and the IRB. The study monitor will also verify that assent was obtained for patients not capable of providing informed consent or that documentation is provided by the investigator explaining why the patient was unable to provide assent. The investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the investigator will permit inspection of the study files by authorized representatives of the regulatory agencies. On completion of the study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

Throughout the course of the study, the medical monitor will determine eligibility of all screened patients, will address any medical issues that might arise, clarify medical questions, review patient safety data (eg, AE/SAE, laboratory, and ECG), and partner with the study team in the overall study management. The study medical monitoring plan will document additional details of the study medical oversight and monitoring.

#### 11 AMENDMENTS

Protocol modifications, except those intended to reduce immediate risk to study patients, may be made only by Boston Pharmaceuticals. A protocol change intended to eliminate an apparent immediate hazard to patients may be implemented immediately, provided the IRB/IEC is notified within 5 days.

Any permanent change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB/IEC and the investigator must await approval before

implementing the changes. Boston Pharmaceuticals will submit protocol amendments to the appropriate regulatory authorities for approval.

If in the judgment of the IRB/IEC, the investigator, and/or Boston Pharmaceuticals, the amendment to the protocol substantially changes the study design and/or increases the potential risk to the patient and/or has an impact on the patient's involvement as a study participant, the currently approved written ICF will require similar modification. In such cases, informed consent will be renewed for patients enrolled in the study before continued participation.

#### 12 STUDY REPORT AND PUBLICATIONS

Boston Pharmaceuticals is responsible for preparing and providing the appropriate regulatory authorities with clinical study reports according to the applicable regulatory requirements.

By signing the protocol, the principal investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the principal investigator's name, address, qualifications, and extent of involvement.

The principal investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted and obtained approval from the sponsor in advance.

#### 13 STUDY DISCONTINUATION

Both Boston Pharmaceuticals and the principal investigator reserve the right to terminate the study at the investigator's site at any time. Should this be necessary, Boston Pharmaceuticals or a specified designee will inform the appropriate regulatory authorities of the termination of the study and the reasons for its termination, and the principal investigator will inform the IRB/IEC of the same. In terminating the study Boston Pharmaceuticals and the principal investigator will assure that adequate consideration is given to the protection of the patients' interests.

#### 14 CONFIDENTIALITY

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from Boston Pharmaceuticals, except to the extent necessary to obtain informed consent from patients who wish to participate in the trial or to comply with regulatory requirements. However, authorized regulatory officials, IRB/IEC personnel, Boston Pharmaceuticals, and its authorized representatives are allowed full access to the records.

Identification of patients and eCRFs shall be by initials, birthdate, or patient number. Documents that identify the patient (eg, the signed informed consent document) must be maintained in confidence by the principal investigator. If required, the patient's full name may be made known to an authorized regulatory agency or other authorized official.

BOS161721


#### 15 REFERENCES

1 Urowitz MB, Gladman DD. How to improve morbidity and mortality in systemic lupus erythematosus. Rheumatology 2000;39:238-44.

- 2 Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, et al. Morbidity and Mortality in Systemic Lupus Erythematosus During a 10-Year Period. Medicine 2003;82(5):299-308.
- 3 Pons-Estel GJ, Alarcón GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010;39(4):257. Epub 2009 Jan 10.
- 4 Kanta H, Mohan C. Three Checkpoints in lupus development: central tolerance in adaptive immunity, peripheral amplification by innate immunity, and end-organ inflammation. Genes and Immunity 2009;10:390-6.
- 5 Dall'Aqua WF, Kiener PA, Wu H. Properties of Human IgG1s Engineered for Enhanced Binding to the Neonatal Fc Receptor (FcRn). J Biol Chem. 2006 Aug 18, 281(33):23514-24.
- 6 Spolski R, Leonard WJ. The Yin and Yang of interleukin-21 in allergy, autoimmunity and cancer. Curr Opin Immunol. 2008a;20:295-301.
- 7 Asao H, Okuyama C, Kumaki S, Ishii N, Tsuchiya S, Foster D, et al. Cutting edge: the common gamma-chain is an indispensable subunit of the IL-21 receptor complex. J Immunol. 2001;167:1-5.
- 8 Habib T, Senadheera S, Weinberg K, Kaushansky K. The common gamma chain (gamma c) is a required signaling component of the IL-21 receptor and supports IL-21-induced cell proliferation via JAK3. Biochemistry. 2002;41:8725-31.
- 9 Spolski R, Leonard WJ. Interleukin-21: basic biology and implications for cancer and autoimmunity. Annu Rev Immunol. 2008b;26:57-79.
- 10 Puga I, Cols M, Barra CM, He B, Cassis L, Gentile M, et al. B-cell-helper neutrophils stimulate the diversification and production of immunoglobulin in the marginal zone of the spleen. Nat Immunol. 2011;13(2):170-80.
- 11 Costanzo A, Chimenti MS, Botti E, Caruso R, Sarra M, Monteleone G. IL-21 in the pathogenesis and treatment of skin diseases. J Dermatol Sci. 2010;60(2):61-6.
- 12 Avery DT, Bryant VL, Ma CS, de Waal Malefy R, Tangye SG. IL-21-induced isotype switching to IgG and IgA by human naive B cells is differentially regulated by IL-4. J Immunol. 2008;181:1767-79.
- 13 Rasmussen TK, Andersen T, Bak, RO, Yiu G, Sorensen CM, Stengaard-Pedersen K, et al. Overexpression of microRNA-155 increases IL-21 mediated STAT3 signaling and IL-21 production in systemic lupus erythematosus. Arthritis Research & Therapy 2015;17(154)


- 14 Ettinger R, Kuchen S, Lipsky PE. The role of IL-21 in regulating B-cell function in health and disease. Immunol Rev. 2008;223:60-86.
- 15 Caprioli F, Sarra M, Caruso R, Stolfi C, Fina D, Sica G, et al. Autocrine regulation of IL-21 production in human T lymphocytes. J Immunol. 2008;180(3):1800-7.
- 16 Yang L, Anderson DE, Baecher-Allan C, Hastings WD, Bettelli E, Oukka M, et al. IL-21 and TGF-beta are required for differentiation of human T(H)17 cells. Nature. 2008;454(7202):350-2.
- 17 Tangye SG, Ma CS, Brink R, Deenick EK. The good, the bad and the ugly TFH cells in human health and disease. Nat Rev Immunol. 2013;13(6):412-26.
- 18 Fantini MC, Rizzo A, Fina D, Caruso R, Becker C, Neurath MF, et al. IL-21 regulates experimental colitis by modulating the balance between Treg and Th17 cells. Eur J Immunol. 2007;37(11):3155-63.
- 19 Peluso I, Fantini MC, Fina D, Caruso R, Boirivant M, MacDonald TT, et al. IL-21 counteracts the regulatory T-cell-mediated suppression of human CD4+ T lymphocytes. J Immunol. 2007;178(2):732-9.
- 20 Hippen KL, Bucher C, Schirm DK, Bearl AM, Brender T, Mink KA, et al. Blocking IL-21 signaling ameliorates xenogeneic GVHD induced by human lymphocytes. Blood. 2012;119(2):619-28.
- 21 Davis ID, Skrumsager BK, Cebon J, Nicholaou T, Barlow JW, Moller NP, et al. An open-label, two-arm, phase I trial of recombinant human interleukin-21 in patients with metastatic melanoma. Clin Cancer Res. 2007;13:3630-6.
- 22 Frederiksen KS, Lundsgaard D, Freeman JA, Hughes SD, Holm TL, Skrumsager BK, et al. IL-21 induces in vivo immune activation of NK cells and CD8(+) T-cells in patients with metastatic melanoma and renal cell carcinoma. Cancer Immunol Immunother. 2008;57(10):1439-49.
- 23 Karrich JJ, Jachimowski LC, Nagasawa M, Kamp A, Balzarolo M, Wolkers MC, et al. IL-21- stimulated human plasmacytoid dendritic cells secrete granzyme B, which impairs their capacity to induce T-cell proliferation. Blood. 2013;121(16):3103-11.
- 24 Lindner S, Dahlke K, Sontheimer K, Hagn M, Kaltenmeier C, Barth TF, et al. Interleukin-21-induced granzyme B-expressing B-cells infiltrate tumors and regulate T-cells. Cancer Res. 2013;73(8):2468-79.
- 25 Monteleone G, Caruso R, Fina D, Peluso I, Gioia V, Stolfi C, et al. Control of matrix metalloproteinase production in human intestinal fibroblasts by interleukin 21. Gut. 2006;55(12):1774-80.
- 26 Nakou M, Papadimitraki ED, Fanouriakis A, Bertsias GK, Choulaki C, Goulidaki N, et al. Interleukin-21 is increased in active systemic lupus erythematosus patients and contributes to the generation of plasma B-cells. Clin Exp Rheumatol. 2013;31(2):172-9.

- 27 Li Q, Liu Z, Dang E, Jin L, He Z, Yang L, et al. Follicular helper T-cells (Tfh) and IL-21 involvement in the pathogenesis of bullous pemphigoid. PLoS One. 2013;8(7):e68145.
- 28 Liu R, Wu Q, Su D, Che N, Chen H, Geng L, et al. A regulatory effect of IL-21 on T follicular helper-like cell and B-cell in rheumatoid arthritis. Arthritis Res Ther. 2012;14(6):R255.
- 29 Kang KY, Kim HO, Kwok SK, Ju JH, Park KS, Sun DI, et al. Impact of interleukin-21 in the pathogenesis of primary Sjögren's syndrome: increased serum levels of interleukin-21 and its expression in the labial salivary glands. Arthritis Res Ther. 2011;13(5):R179.
- 30 Terrier B, Geri G, Chaara W, Allenbach Y, Rosenzwajg M, Costedoat-Chalumeau N, et al. Interleukin-21 modulates Th1 and Th17 responses in gianT-cell arteritis. Arthritis Rheum. 2012a;64(6):2001-11.
- 31 Terrier B, Costedoat-Chalumeau N, Garrido M, Geri G, Rosenzwajg M, Musset L, et al. Interleukin 21 correlates with T-cell and B-cell subset alterations in systemic lupus erythematosus. J Rheumatol. 2012b;39(9):1819-28.
- 32 International Conference on Harmonisation. Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals S6 (R1). 2011.
- 33 Wang W, Wang EQ, Balthasar JP. Monoclonal Antibody Pharmacokinetics and Pharmacodynamics. Clin Pharm & Ther 2008; 84(5):548-58.
- 34 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 35 Elsaesser H, Sauer K, Brooks DG. IL-21 is required to control chronic viral infection. Science. 2009;324(5934):1569-72
- 36 Kotlarz D, Zietara N, Uzel G, Weidemann T, Braun CJ, Diestelhorst J, et al. Loss-of-function mutations in the IL-21 receptor gene cause a primary immunodeficiency syndrome. J Exp Med. 2013;210(3):433-43.
- 37 Hunter PR, Nichols G. Epidemiology and clinical features of Cryptosporidium infection in immunocompromised patients. Clinical microbiology reviews. 2002;15(1):145-54.
- 38 Desjardins M, Mazer BD. B-cell memory and primary immune deficiencies: interleukin-21 related defects. Curr Opin Allergy Clin Immunol. 2013;13(6):639-45.
- 39 Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. *Nephron*. 1976;16(1):31-41.
- 40 Guidelines for Using the QuantiFERON®-TB Gold Test for Detecting Mycobacterium tuberculosis Infection, US: http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5415a4.htm.

41 NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, available at https://evs.nci.nih.gov/ftp1/CTCAE/About.html.

- 42 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 43 Posner K, Melvin G a, Stanley B, Oquendo M a, Gould M. Factors in the assessment of suicidality in youth. *CNS Spectr*. 2007;12(2):156-162.
- 44 Castrejon I, Tani C, Jolly M, Huang A, Mosca M. Indices to assess patients with systemic lupus erythematosus in clinical trials, long-term observational studies, and clinical care. Clin Exp Rheumatol 2014; 32(85):S85-95.
- 45 Furie R, Wang L, Drappa J, Illei G. Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] Response Is Associated with Global Benefit in Patients with Moderate to Severe SLE [abstract]. *Arthritis Rheumatol.* 2016; 68 (suppl 10).
- 46 Thanou A, Chakravarty E, James JA, Merrill JT. Which outcome measures in SLE clinical trials best reflect medical judgment? Lupus Science & Medicine 2014;1:e000005. doi:10.1136/lupus-2013-000005.
- 47 Wallace DJ, Kalunian K, Petri MA, Strand V, Houssiau FA, Pike M, et al. Efficacy and safety of epratuzumab in patients with moderate/severe active systemic lupus erythematosus: results from EMBLEM, a phase IIb, randomised, double-blind, placebo-controlled, multicentre study. *Ann Rheum Dis* 2014;73:183-90.
- 48 Albrecht J, Taylor L, Berlin JA, Dulay S, Ang G, Fakharzadeh S. The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index): An Outcome Instrument for Cutaneous Lupus Erythematosus. J Invest Derm. 2005;125(5):889-94.
- 49 Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is Valid, and Renal and Pulmonary Organ Scores are Predictors of Sever Outcome in Patients with Systemic Lupus Erythematosus. Br J Rheumatol. 1996;35:248-54.



# 16 APPENDICES

# APPENDIX 1 NAMES OF STUDY PERSONNEL

Sponsor: Boston Pharmaceuticals
55 Cambridge Parkway Suite 401
Cambridge, MA 02142, USA

Medical Monitor:

PPD

Clinical Research
Organizations:

PPD

PPD

Bioanalytical Laboratory:

PPD

Central Laboratory:

PPD


# APPENDIX 2 DECLARATION OF HELSINKI

#### WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI

Ethical Principles
For
Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly
Helsinki, Finland, June 1964
and amended by the
29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
and the

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### A. INTRODUCTION

The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.

It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.

The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my subject will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the subject's interest when providing medical care which might have the effect of weakening the physical and mental condition of the subject."

Medical progress is based on research, which ultimately must rest in part on experimentation involving human subjects.

In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.

The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic, and therapeutic procedures and the understanding of the etiology and pathogenesis of disease. Even the best-proven prophylactic, diagnostic, and therapeutic methods must continuously be challenged through research for their effectiveness, efficiency, accessibility, and quality.

In current medical practice and in medical research, most prophylactic, diagnostic, and

therapeutic procedures involve risks and burdens.

Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.

Research investigators should be aware of the ethical, legal, and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal, or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### В. BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.

Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.

Appropriate caution must be exercised in the conduct of research, which may affect the environment, and the welfare of animals used for research must be respected.

The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any SAEs. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.

The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles enunciated in this Declaration.

Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a subject of the research, even though the subject has given consent.

Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the

subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.

Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.

Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.

Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.

The subjects must be volunteers and informed participants in the research project.

The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the subject's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.

In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.

When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.

For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the investigator must obtain informed consent from the legally authorized representative in accordance with applicable law. These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.

When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the investigator must obtain that assent in addition to the consent of the legally authorized representative.

Research on individuals from whom it is not possible to obtain consent, including proxy or advance consent, should be done only if the physical/mental condition that prevents obtaining

informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.

Both authors and publishers have ethical obligations. In publication of the results of research, the investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic, or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the subjects who are research subjects.

The benefits, risks, burdens, and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic, or therapeutic method exists.

At the conclusion of the study, every subject entered into the study should be assured of access to the best-proven prophylactic, diagnostic, and therapeutic methods identified by the study.

The physician should fully inform the subject which aspects of the care are related to the research. The refusal of a subject to participate in a study must never interfere with the subject-physician relationship.

In the treatment of a subject, where proven prophylactic, diagnostic, and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the subject, must be free to use unproven or new prophylactic, diagnostic, and therapeutic measures, if in the physician's judgment it offers hope of saving life, re-establishing health, or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases, new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.

BOS161721 Boston Pharmaceuticals, Inc.


# APPENDIX 3 COMMONLY USED CORTICOSTEROID EQUIVALENTS

| Medication | Dose Equivalence |
|--------------------|------------------|
| Prednisone | 20 mg |
| Cortisone | 100 mg |
| Hydrocortisone | 80 mg |
| Prednisolone | 20 mg |
| Methylprednisolone | 16 mg |
| Triamcinolone | 16 mg |
| Budesonide | 4 mg |
| Dexamethasone | 3 mg |
| Bethamethasone | 2.4 mg |

# APPENDIX 4 MEDICATION WASHOUT PERIODS

# WASHOUT TIMES OF MEDICATIONS BASED ON 5 HALF-LIVES

| Medication | Discontinuing Prior to Signing Consent |
|---|---|
| Abatacept (CTLA4Ig) | 24 weeks |
| Alefacept | 12 weeks |
| AMG 623 (blisibimod) | 24 weeks |
| Anifrolumab | 12 weeks |
| Atacicept (TACI-Ig) | 12 weeks |
| Belimumab | 24 weeks |
| Cyclophosphamide | 24 weeks |
| Cyclosporine (except for CSA eye drops) | 4 weeks |
| Danazol | 4 weeks |
| Dapsone | 4 weeks |
| Eculizumab | 12 weeks |
| Efalizumab | 12 weeks |
| Epratuzumab | 24 weeks |
| Intravenous globulin | 4 weeks |
| Leflunomide | 8 weeks (4 weeks for washout with |
| | cholestyramine) |
| Lenalidomide with cholestiramine | 8 weeks |
| Lupuzor | 12 weeks |
| Memantine | 4 weeks |
| Natalizumab | 24 weeks |
| Ocrelizumab | 48 weeks (or 24 weeks with recovery of B cell) |
| Pimecrolimus | 4 weeks |
| Plasmapheresis | 24 weeks |
| Retinoids (oral or topical) | 4 weeks |
| Rituximab | 48 weeks (or 24 weeks with recovery of B cell) |
| Sirolimus | 4 weeks |
| Tacrolimus | 4 weeks |
| Thalidomide | 8 weeks |
| Tocilizumab | 12 weeks |

# APPENDIX 5 BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA)



# APPENDIX 6 INJECTION SITE REACTION GRADING SCALE

| Adverse event Injection site reaction | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Definition: A disorder<br>characterized by an<br>intense adverse reaction<br>(usually immunologic)<br>developing at the site of<br>an injection | Tenderness with or without associated symptoms (eg, warmth, erythema, itching) | Pain;<br>Lipodystrophy;<br>Edema;<br>phlebitis | Ulceration or<br>necrosis;<br>Severe tissue<br>damage;<br>Operative<br>intervention<br>indicated | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>indicated | Death |
| Pain | Mild pain | Moderate pain;<br>limiting<br>instrumental ADL | Severe pain;<br>limiting self-<br>care ADL | - | - |
| Rash<br>maculopapular/Erythem<br>a/Induration | Macules/papules<br>covering <10%<br>BSA with or<br>without | Macules/papules<br>covering 10% - 30%<br>BSA with or<br>without symptoms | Macules/papul<br>es covering<br>> 30% BSA<br>with or | - | - |
| Definition: A disorder characterized by the presence of macules (flat) and papules (elevated). Also known as morbillform rash, it is | symptoms (eg, pruritus, burning, tightness) Erythema covering <10% | (eg, pruritus,<br>burning, tightness);<br>limiting<br>instrumental ADL;<br>Erythema 30% BSA<br>with or without | without<br>associated<br>symptoms;<br>limiting<br>self-care ADL | | |
| one of the most<br>common cutaneous<br>adverse events,<br>frequently affecting the<br>upper trunk, spreading<br>centripetally, and | BSA with or without symptoms (eg, pruritus, burning, tightness) | symptoms (eg,<br>pruritus, burning,<br>tightness); limiting<br>instrumental ADL | Erythema covering > 30% BSA with or without associated | | |
| associated with pruritus. | | | symptoms;<br>limiting<br>self-careADL | | |

ADL = active daily living

# APPENDIX 7 PROTOCOL SUMMARY OF CHANGES

The protocol summary of changes was moved to the end of the protocol for easier readability.

Significant changes are described in the table below. Changed text is displayed for the first major occurrence only. Deleted text is presented in strikethrough format, and added text is presented in bold format.

| Section | Description of Changes | Rationale |
|---|---|---|
| Global | Add: | Administrative |
| | Added 'Protocol Date and Version: 21 March 2018; V3.0' to the header. | |
| Global | Change: | Administrative |
| | Changed Version number from V2.0 (Amendment 1) to V3.0 (Amendment 2) and Version date from 14 November 2017 to 21 March 2018. | |
| Global | Change: | Replaced |
| | Changed subjects to <b>patients</b> . | 'subjects' to 'patients' since the enrolled participants are with SLE condition |
| Global | Made administrative and editorial (formatting, typographical, and grammatical) updates. | Administrative |
| PROTOCOL<br>SUMMARY, | Add: | Clarification that POC dose |
| Background and<br>Rationale | The Phase 2 portion will be a proof of concept (POC) study, where dose selection will be based on the <b>data monitoring committee (DMC) and</b> sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD study of 30 patients treated with BOS161721/placebo | selection will<br>be based on<br>DMC and<br>sponsor<br>assessment |
| PROTOCOL<br>SUMMARY,<br>Objectives and<br>Endpoints | The objectives and endpoints sections were combined together and are now represented in a table format in order to demonstrate which endpoints correspond to each objective. Only primary and secondary objectives and endpoints are listed within the synopsis. Additional edits were made to some objectives and endpoints. Some new endpoints were added to the study. | Updated for<br>clarity and to<br>provide a<br>comprehensive<br>list of<br>endpoints<br>identified in |
| | An exploratory objective, to examine PK and PD effects of BOS161721 in subjects with mild to moderate SLE, was changed to 'secondary objective'. | the protocol |
| | Changes to the objectives and endpoints are noted below: | |
| | MAD Phase 1b Study | |

# Section Description of Changes

Rationale

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose. | Safety Endpoints Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness Injection site reactions Columbia Suicide severity Rating Scale (C-SSRS) 12-lead electrocardiograms (ECGs) parameter results at each visit and change from baseline Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline Clinical laboratory results and change from baseline Clinical examinations changes from baseline Anti-drug antibodies (ADAs) Study drug exposure/compliance |
| | Concomitant medication |
| Secondary | usage |
| To characterize the PK of<br>BOS161721 and select the<br>optimal dose of BOS161721<br>based on safety, PK, and PD<br>effects in patients with mild to<br>moderate SLE. | <ul> <li>Pharmacokinetic Endpoints</li> <li>BOS161721 concentration by visit and time point</li> <li>Maximum observed concentration (C<sub>max</sub>), first time to maximum concentration (T<sub>max</sub>), area under the concentration-time curve (AUC), t<sub>1/2</sub>, systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>)</li> </ul> |
| | Pharmacodynamic Endpoints Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype Results and changes (or shifts) from baseline in anti-double-stranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B |

# Section Description of Changes

#### Rationale



The rules for CS usage during the trial, as well as limitations of other prohibited medications, are applied on the analytical end to ensure SRI-4 responders meet all necessary criteria.
# Section Description of Changes

Rationale



# **POC Phase 2 Study**

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To demonstrate a superior effect of<br>BOS161721 at the chosen dose<br>compared with placebo for response<br>on the SLE Responder Index 4<br>(SRI-4) | • The proportion of subjects with a SRI-4 response at Day 210 (see Section 6.3.4.1) |
| Secondary | |

# Section Description of Changes

Rationale

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment

## Secondary Efficacy Endpoints

- The proportion of subjects with:
  - SRI-4 response at each visit
  - SRI-5 and SRI-6 response (Section 6.3.4.2)
  - a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210
  - new BILAG A flare or > 1 BILAG B flares relative to baseline through Day 210
  - PGA worsening
  - a BICLA response
  - a CLASI response
  - medication failures
- Results and changes from baseline in:
  - CLASI
  - swollen and tender joints ACR-28
  - SLEDAI-2K
  - SLICC/ACR damage index
- Time to medication failure
- Duration of SRI-4 response
- Time to first SRI-4 response
- Time to BILAG A flare or
   1 BILAG B flare
   compared to baseline
   through Day 210

#### Safety

 To assess safety and tolerability of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment

#### **Safety Endpoints**

- Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness
- Injection site reactions
- C-SSRS
- 12-lead ECGs parameter results at each visit and change from baseline
- Vital signs (blood

Section Description of Changes Rationale




#### Section **Description of Changes** Rationale **PROTOCOL** Replace: Clarification that patients SUMMARY, Study Design The trial will consist of a staggered MAD Phase 1b and POC Phase 2 will not have studies. Both studies will be double blinded with each patient having the the same same number of doses (7), and visits; the duration will be 180 days, number of followed by a 90-day follow-up safety observation period. visits in both studies. With: The trial will consist of 2 double-blinded studies: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270. Delete: The futility **PROTOCOL** analysis was SUMMARY, removed due Study Design Two weeks after the last patient in Cohort 3 receives the second dose, the DMC and Boston Pharmaceuticals will conduct a data review for the first to the modest size of the trial Section 1.2.4, interim analysis (IA1). At that time, a decision will be made to suggest but more Risk-Benefit which dose should be carried forward into the POC Phase 2 study. importantly Assessment because the least reliable data (high placebo response) is known to occur during the first half of the study (before week 24) when futility analysis was planned **PROTOCOL** Add: Clarification SUMMARY, on POC Study Design sample size For the POC study, approximately 156 additional patients will be randomized to active or placebo groups in a 2:1 ratio. Section 3.1.2.2, POC Study Design

BOS161721 Boston Pharmaceuticals, Inc.


#### Section

## **Description of Changes**

# PROTOCOL SUMMARY, Study Design

# Replace:

Data from 60 patients, including the 12 from the MAD study, or 6 fewer if the low dose is chosen, who are in the cohort of the chosen dose for the POC study who complete 3 months of treatment will be used in a second IA (IA2) at Day 90 to assess if the trial could stop for an early futility conclusion. If futility is not claimed in the IA2, the POC study will continue to approximately 156 patients.

Following the 6 month treatment period, primary and secondary efficacy endpoints will be assessed for each patient, after providing their Day 180 disease activity assessments. DMC monitoring will be conducted periodically throughout the study as described in the DMC charter.

## With:

DMC **safety reviews** will be conducted periodically throughout the study as described in the DMC charter.

# Rationale

Removed assessment information from section, and the futility analysis was removed due to the modest size of the trial but more importantly because the least reliable data (high placebo response) is known to occur during the first half of the study (before week 24) when FA was planned

# PROTOCOL SUMMARY,

Main Criteria for Inclusion and Exclusion (inclusion criterion 6, subbullet ii)

Section 4.4, Inclusion Criteria (inclusion criterion 6,

sub-bullet ii)

# Replace:

ii Points from lupus headache and organic brain syndrome are also excluded

#### With:

ii Points from lupus headache and organic brain syndrome will also be excluded

Corrected to maintain consistency

#### Section

# **Description of Changes**

## PROTOCOL SUMMARY,

Main Criteria for Inclusion and Exclusion (inclusion criterion 7, subbullets a and b)

#### Replace:

- 7 Patients must have at least 1 of the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 4.4.
  - c If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

With:

- 7 Patients must have at least 1**A or 2Bs from** the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a BILAG A or B score in the mucocutaneous body system
  - b BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 4.4.

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores

# PROTOCOL SUMMARY,

Statistical Considerations

#### Replace:

Baseline and patient characteristics will be summarized via appropriate summary statistics by treatment group and overall, for each phase of the trial.

Binary efficacy endpoints will be compared between treatments via Cochran-Mantel-Haenszel (CMH) analysis. Continuous efficacy endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-by-time interaction, baseline covariate, and covariate-by-time interaction. Summary statistics will be provided by dose/treatment for all safety endpoints. Details will be provided in the statistical analysis plan (SAP).

Two IAs are planned for this study. The initial IA (IA1) will be conducted at the time of the POC decision for dose selection. The second IA (IA2)

#### Rationale

Text updated to clarify that a minimum BILAG 1 'A' or 2 'B' scores is required for screening

The futility analysis was removed due to the modest size of the trial but more importantly because the least reliable data (high placebo response) is known to occur during the first half of the study (before week

#### Section

## **Description of Changes**

will be performed for futility. IA2 is planned to be conducted when SRI-4 response is determined for approximately 60 patients (including all patients at the same dose level/matching placebo from the MAD study) after completing 3 months of treatment. The purpose of IA2 is to assess if the trial could stop for an early futility conclusion, or continue. Since there is no plan to stop the trial for an early efficacy conclusion, there is no impact on the type 1 error level.

AEs will be summarized by counts and percentages of patients by treatment group. Laboratory data and vital signs will be summarized by treatment group as summary statistics for value and change from baseline at each individual time point. Summary statistics will include n, arithmetic mean, median, arithmetic SD, minimum, and maximum.

The PK parameter data will be listed and summarized descriptively in tabular format. Binary PD endpoints will be assessed for the full analysis set (FAS) population via CMH analysis. Continuous PD endpoints will be assessed via ANCOVA repeated measures mixed model analysis with multiple factors. PK and PD relationships will be explored graphically and where appropriate model based methods of analysis will used.

#### With:

Two analyses are planned: 1) an interim analysis to select the Phase 2 dose based on Phase 1 data, and 2) a final analysis at study completion. Additionally, DMC safety analyses will be performed after each Phase 1 cohort and throughout Phase 2 to monitor patient safety.

Unless stated otherwise, statistical testing will only be performed on the Phase 2 data and will be done using 2-sided overall alpha of 0.10. Data will be summarized descriptively by treatment and overall for each study phase. For the MAD phase, BOS161721 will be summarized overall and by each dose level and placebo patients from each cohort will be combined.

The descriptive summaries for the categorical data will include number and percentage. The descriptive summaries for the continuous data will include number, mean, standard deviations (SD), 25th and 75th percentiles, minimum, median, and maximum. Counts medians, 25th and 75th percentiles, and standard error will be presented for time-to-event data.

All safety analyses will be performed using the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. All efficacy analyses will be performed using the full analysis set (FAS), defined as all patients who have receive at least 1 dose of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. Select efficacy analyses may also be performed on the per protocol (PP) set.

Binary efficacy endpoints, including the primary efficacy endpoint, will

#### Rationale

24) when futility analysis was planned

Text updated to allow use of testing procedures that are not typical/straight forward as 1-sided (such as CMH).

Simplification and consistency with binary endpoints. Allows more

## Section Description of Changes

BOS161721

#### Rationale

be assessed via Pearson's chi-squared analysis.

flexibility in handling missing data.

Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) when applicable, adjusting for the baseline value. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test.

Adverse event data will be coded to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class and preferred term will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be summarized, based on coded terms, using frequency and percentage of patients. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters, will be summarized at each individual visit.

# List of Abbreviations

Add:

ANOVA analysis of variance ANCOVA analysis of covariance CS corticosteroids

CCI

FAS full analysis set

MedDRA Medical Dictionary of Regulatory Activities PP per protocol

safety analysis set

SS Delete:

List of Abbreviations

RNP ribonucleoprotein

Updated to align with abbreviations deleted throughout the

protocol

Updated to

align with abbreviations

throughout the

added

protocol

## Section 1.2.3, Study Dose Selection

Delete:

In addition, the DMC and Boston Pharmaceuticals will conduct a data review—for the first interim analysis (IA1). At that time, a decision will be made to suggest which dose should be carried forward into the proof of concept (POC) Phase 2 study.

The futility analysis was removed due to the modest size of the trial but more importantly Clinical Study Protocol: BOS161721-02


# Section Description of Changes Rationale

because the least reliable data (high placebo response) is known to occur during the first half of the study (before week 24) when futility analysis was planned

Section 1.2.4, Risk-Benefit Assessment Replace:

Thereafter, DMC monitoring will be conducted periodically throughout the study as described in the DMC charter.

With:

Thereafter, DMC **safety reviews** will be conducted periodically throughout the study as described in the DMC charter.

for clarification

Text updated


# Protocol Date and Version: 21 March 2018; V3.0 Section Description of Changes

# Section 2, Study Objectives And Endpoints

Replace:

This trial has separate primary and secondary objectives for the MAD Phase 1b and POC Phase 2 studies.

Text updated to appropriately setup table

Rationale

#### With:

This trial has separate objectives and endpoints for the MAD Phase 1b and POC Phase 2 studies. The primary, secondary, and exploratory objectives for each phase, as applicable, are described below with their corresponding endpoints.

# Section 2, Study Objectives And Endpoints

The objectives and endpoints sections (Section 2 and 3 in Amendment 1) were combined into 1 section (Section 2 of Amendment 2) and the objectives and endpoints are now in a table format to easily distinguish which endpoints align with each objective. Additional edits were made to the objectives and endpoints. Some new endpoints were added to the study.

An exploratory objective, to examine PK and PD effects of BOS161721 in subjects with mild to moderate SLE, was changed to 'secondary objective'.

Updated for clarity and to provide a comprehensive list of endpoints identified in the protocol

Changes to the objectives and endpoints are noted below:

#### 2.1 Phase 1b Multiple Ascending Dose

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose. | Safety Endpoints Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness Injection site reactions Columbia Suicide severity Rating Scale (C-SSRS) 12-lead electrocardiograms (ECGs) parameter results at each visit and change from baseline Vital signs (blood pressure [BP], heart rate, and temperature) parameter results at each visit and change from baseline Clinical laboratory results and change from baseline Physical examinations changes from baseline ADAs Study drug |


#### Section **Description of Changes**

Rationale

# exposure/compliance Concomitant medication usage Secondary To characterize the PK of **Pharmacokinetic Endpoints** BOS161721 and select the BOS161721 concentration by optimal dose of BOS161721 visit and time point based on safety, PK, and PD Maximum observed effects in patients with mild to concentration ( $C_{max}$ ), $T_{max}$ , area moderate SLE. under the concentration-time curve (AUC), terminal elimination half-life (t1/4) systematic clearance (C<sub>L</sub>), volume of distribution (V<sub>d</sub>) **Pharmacodynamic Endpoints** Results and changes (or shifts) from baseline to each visit in phosphorylated signal transducer and activator of transcription 3 (pSTAT3), C3 and C4 levels, and leukocyte immunophenotype Results and changes (or shifts) from baseline in anti-doublestranded DNA (dsDNA), antinuclear antibodies (ANA), anti-Sjögren syndrome A and B (SSA, SSB), Smith (Sm), and antiphospholipid (APL) autoantibodies at each visit Results and changes (or shifts) from baseline in abrogation of IL-21 gene signature at each indicated visit **Exploratory**

# Section Description of Changes

Rationale



# 2.2 Phase 2 Proof of Concept

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To demonstrate a superior effect of<br>BOS161721 at the chosen dose<br>compared with placebo for response<br>on the SLE Responder Index 4<br>(SRI-4) | <ul> <li>Primary Efficacy Endpoint</li> <li>The proportion of subjects with a SRI-4 response at Day 210 (see Section 6.3.4.1)</li> </ul> |
| Secondary | |

The rules for CS usage during the trial, as well as limitations of other prohibited medications, are applied on

# Section Description of Changes

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment

# Secondary Efficacy Endpoints

- The proportion of subjects with:
  - SRI-4 response at each visit
  - SRI-5 and SRI-6 response (Section 6.3.4.2)
  - a sustained reduction of oral corticosteroid (CS) (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210
  - new BILAG A flare or > 1 BILAG B flares relative to baseline through Day 210
  - PGA worsening
  - a BICLA response
  - a CLASI response
  - medication failures
- Results and changes from baseline in:
  - CLASI
  - swollen and tender joints ACR-28
  - SLEDAI-2K
  - SLICC/ACR damage index
- Time to medication failure
- Duration of SRI-4 response
- Time to first SRI-4 response
- Time to BILAG A flare or
   1 BILAG B flare
   compared to baseline
   through Day 210

## Rationale

the analytical end to ensure SRI-4 responders meet all necessary criteria.

#### Safety

 To assess safety and tolerability of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment

#### **Safety Endpoints**

- Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), related AEs, AEs leading to study drug discontinuation, AEs by severity and relatedness
- Injection site reactions
- C-SSRS
- 12-lead ECGs parameter results at each visit and change from baseline
- Vital signs (blood pressure

# Section Description of Changes

## Rationale



Section 3.1, Study Design

Replace:

The trial will consist of 2 studies: MAD Phase 1b, and POC Phase 2. Both studies will be double-blinded, and patients will have the same number of visits. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by a 90-day safety follow-up visit.

Text updated to correspond with POC portion having 1 less visit.


rotocol Date and Version: 21 March 2018;

# Section Description of Changes

Rationale

With:

The trial will consist of 2 **double-blinded** studies: MAD Phase 1b and POC Phase 2. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by **safety follow-up visits at Days 210, 240, and 270.** 

Section 3.1.1.1,

Dose Escalation for the MAD Study

Replace:

If > 3 patients discontinue the study in a cohort, he/she may be replaced.

With:

If patients discontinue the study in a cohort **prior to adequate safety follow-up**, he/she may be replaced.

to clarify that replacement may occur if any amount of subjects discontinue too early to establish safety

Updated text

Section 3.1.1.3,

DMC

Recommendations

Delete:

For the POC study, the DMC and Boston Pharmaceuticals will conduct a data review for the IA1 to suggest which dose should be carried forward into the POC Phase 2 study.

The futility analysis was removed due to the modest size of the trial but more importantly because the least reliable data (high placebo response) is known to occur during the first half of the study (before week 24) when FA was planned.

Section 3.1.2.2,

POC Study

Design

Add:

Dose selection will be based on the **DMC and** sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD study of 30 patients treated with BOS161721/placebo.

Clarification that POC dose selection will be based on DMC and sponsor assessment

Section 3.1.2.2,

POC Study Design Replace:

Data from approximately 60 patients (including the 12 from the MAD study, or 6 fewer if the low dose is chosen who are in the cohort of the chosen dose for the POC study) who complete 3 months of treatment will be used in the IA2 at Day 90 to assess if the trial could stop for an early futility conclusion (see Section 9.3 for details regarding the IA). If futility is not claimed in the IA2, the POC study will continue to approximately

Removed assessment information from section and the futility analysis was removed due to the modest

#### Section

## **Description of Changes**

156 patients.

Following the 6-month treatment period, primary and secondary efficacy endpoints will be assessed for each patient after providing their Day 180 disease activity assessments.

DMC monitoring will be conducted periodically throughout the study as described in the DMC charter.

With:

DMC **safety reviews** will be conducted periodically throughout the study as described in the DMC charter.

# Section 3.2, Randomization and Blinding (new section)

#### Add:

#### 3.2 Randomization and Blinding

This is a randomized, double-blind study.

Patients meeting all inclusion and exclusion criteria will be centrally randomized to either placebo or BOS161721 using an IWRS according to a randomization list generated by an independent, non-study statistician. Randomization will be performed separately for each study phase and separately for each cohort in the Phase 1b and 2 portion as follows:

| Phase/Cohort | Number of Patients | Randomization Ratio<br>BOS161721:Placebo |
|---|---|---|
| Phase<br>1b/Cohort 1 | 6 | 5:1 |
| Phase<br>1b/Cohort 2 | 12 | 3:1 |
| Phase<br>1b/Cohort 3 | 12 | 3:1 |
| Phase 2 | 156* | 2:1 |

\*Additional patients may be enrolled to confirm sufficient numbers of patients are in the full analysis set (FAS).

Eligible patients will be assigned to the study phase which is active at time of enrollment. Similarly, patients in the Phase 1 MAD will be assigned to the cohort which is active. Each patient will be assigned a unique randomization number which will not be reused.

All patients, investigators, and study team participants will be blinded to treatment assignment. An independent biostatistician not otherwise involved on the study will be unblinded and prepare materials for the interim analysis (IA) and the DMC safety reviews.

#### Rationale

size of the trial but more importantly because the least reliable data (high placebo response) is known to occur during the first half of the study (before week 24) when FA was planned

Text was added to clarify randomization and blinding process

## Section

## **Description of Changes**

Rationale

The DMC will review unblinded data during safety reviews and the IA. A limited team at Boston Pharmaceuticals will review unblinded results from the Phase 1b MAD portion during the IA to determine the dose that will be used for the Phase 2 POC portion of the study. Details regarding maintenance of the blinding and content of data reviews will be described in the DMC charter or related study documentation.

# Section 3.3, Study Schematic

## Replace:



The futility analysis was removed due to the modest size of the trial but more importantly because the least reliable data (high placebo response) is known to occur during the first half of the study (before week 24) when futility analysis was planned

## With:



Section 3.4, Schedule of Assessments (Table 1)

# Replace:

| | Screen <sup>a</sup> | Enroll | Treatment Period<br>Follow-Up | | |
|---|---|---|---|---|---|
| | -28 | | 7 15 30 | | |
| Days | to -1 | 0 | (± 1) | $(\pm 3)$ | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 |
| Injection site reaction assessment <sup>f</sup> | | X | X | | X |
| Plasma CCI & | X | X | | X | X |
| Whole blood for | X | X | | X | X |

Clarification of when certain assessments will be collected

# Section Description of Changes Rationale

| leukocyte<br>immunophenotype | | | | |
|------------------------------|---|---|---|---|
| CCI | | X | X | X |
| CCI | | | | |
| | X | X | | X |

# With:

| | Screen <sup>a</sup> | Enroll | | Treatment Pe<br>Follow-U | |
|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 |
| Injection site reaction assessment | | X <sup>f</sup> | X | | X |
| Plasma CCI & | | X | | X | X |
| Whole blood for leukocyte | | | | | |
| immunophenotype | | X | | X | X |
| CCI | | X | | X | |
| CCI | | | | | |
| | X | X | | | X |


## Section

## **Description of Changes**

# Section 3.4, Schedule of Assessments (Table 1)

#### Replace:

| | Treatmer | nt Period F | ollow-Up | Safe | ety Follow- | -up |
|--------|----------|-------------|----------|-------|-------------|-------|
| | 150 | 180 | 187 | 195 | 210 | 240 |
| Days | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit | | | | | | |
| number | 9 | 10 | | | 11 | 12 |
| pSTAT3 | X | | | | | X |

## Rationale

Clarification of when certain assessments will be collected

With:

| | Treatment Period Follow-Up Safety Follow-up | | | -up | | |
|---|---|---|---|---|---|---|
| | 150 | 180 | 187 | 195 | 210 | 240 |
| Days | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit number | 9 | 10 | | | 11 | 12 |
| pSTAT3 <sup>1</sup> | | | | | | |

Section 3.4, Schedule of Assessments (Table 1 footnotes) Add:

- i When clinically indicated for hemolytic anemia.
- 1 Predose (trough) samples only.

# Section 3.4, Schedule of Assessments (Table 1 and its footnotes)

Delete:

- Predose<sup>e</sup>
- f Injection site reaction assessments to be performed predose and at 2 hours postdose.
- o Predose samples occur on study drug administration visit days.

Text added to maintain consistency throughout the document.

Clarified that no need for predose injection site reaction assessment at baseline and definition of 'o' was deleted as it was redundant.

Clarification of when certain assessments will be collected

Section 3.4, Schedule of Assessments (Table 2)

## Replace:

| | Screen <sup>a</sup> | Enroll | Treatment Period<br>Follow-Up | | |
|---|---|---|---|---|---|
| | -28 | | 15 | 15 30 60 | |
| Days | to -1 | 0 | $(\pm 3)$ | $(\pm 3)$ | $(\pm 3)$ |
| Visit Number | 1 | 2 | 3 | 4 | 5 |
| Injection site reaction assessment <sup>f</sup> | | X | | X | X |
| Plasma CC & | X | X | X | X | X |
| Whole blood for leukocyte immunophenotype | X | X | X | X | X |

## Section

# **Description of Changes**

Rationale

| CCI | | X | X | X | |
|-----|---|---|---|---|---|
| CCI | | | | | |
| | X | X | | X | X |

With:

| | Screen <sup>a</sup> | Enroll | Treatment Period<br>Follow-Up | | |
|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 |
| Injection site reaction assessment | | X <sup>f</sup> | | X | X |
| Plasma CCI & | | X | X | X | |
| Whole blood for leukocyte immunophenotype | | X | X | X | |
| CCI | | X | X | | |
| CCI | X | X | | X | X |

Section 3.4, Schedule of Assessments (Table 2 footnotes) Add:

When clinically indicated for hemolytic anemia.

Section 3.4, Schedule of Assessments (Table 2 footnotes) Delete:

pSTAT3<sup>1</sup>Predose<sup>q</sup>

f Injection site reaction assessments to be performed predose and at 2 hours postdose.

l Predose (trough) samples only.

q Predose samples occur on study drug administration visit days.

Text added to maintain consistency throughout the document.

Clarified that no need for predose injection site reaction assessment at baseline, definition of 'q' was deleted as it was redundant, and footnote 'l' was removed to align with removal of pSTAT3 from the table

Section 4.2, Number of Patients Add:

Approximately 30 patients will be randomized for the MAD Phase 1b study, and approximately 156 **additional** patients will be randomized in

Clarification on POC sample size


#### Section **Description of Changes** Rationale the POC Phase 2 study. Section 4.2, Replace: Text updated Number of to clarify new number of Patients Note that approximately 30 dropouts are assumed. dropouts assumed for With: the study Note that approximately 24 dropouts are assumed. Section 4.4, Replace: Text updated Inclusion Criteria to clarify that a minimum (Inclusion Patients must have at least 1 of the following manifestations of criterion 7, part b, BILAG 1 'A' SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer: or 2 'B' scores subparts i and ii) is required for BILAG A or B score in the mucocutaneous body system screening

- BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
  - i. "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis in  $\geq 2$  joints with marked loss of functional range of movements and significant impairment of basic activities of daily living that has been present on several days cumulatively over the past 4 weeks, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
    - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):
      - Ambulation, toileting, grooming- including bathing and dressing; feeding oneself, (and not responsive to steroids up to 10 mg/day, antimalarials, NSAIDs)
  - "BILAG B:" Moderate Arthritis, Tendonitis or ii. Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in  $\geq 1$  joint, (observed or throughout history), with some loss of functional range of movements which lead to some loss of functional range of motion as manifested by effects on instrumental ADLs such as:
    - Cooking, driving, using the telephone or computer, shopping, cleaning, etc, and has been present on several days over the last 4 weeks, and is present at the time of the screening visit
- If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body

# Section Description of Changes

Rationale

systems for a total of 2 "B" BILAG body system scores

With:

- 7 Patients must have at least 1A or 2Bs from the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a BILAG A or B score in the mucocutaneous body system
  - b BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - i "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis in ≥ 2 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living that has been present on several days cumulatively over the past 30 days, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
      - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):
        - Ambulation, toileting, grooming- including bathing and dressing; feeding oneself
    - ii "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in ≥ 1 joint, (observed or throughout history), with some loss of functional range of movements which lead to some loss of functional range of motion as manifested by effects on instrumental ADLs such as:
      - Cooking, driving, using the telephone or computer, shopping, cleaning, etc, and has been present on several days over the last 30 days, and is present at the time of the screening visit

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores


#### Section **Description of Changes** Rationale Section 5.1, Add: Text updated to clarity Screening Direct Coomb's test (if indicated for hemolytic anemia) Section 5.2, Enrollment/Rando mization and Day 0 Treatment Section 5.3, Treatment Period/Follow-Up Visits Section 5.4, Safety Follow-Up Visits Section 5.1, Delete: Updated to Screening clarify the planned CD4+ count, total IgG and IgM levels, plasma , <del>plasma</del> whole blood for leukocyte laboratory and CC assessments immunophenotype; CC Section 5.1.1, Add: Text added for Retesting During further Screening Period there is evidence a laboratory sample was mislabeled, indeterminate, clarification inadequately processed, and/or deteriorated in transit to the central laboratory Updated to Section 5.2, Replace: clarify the Enrollment/Rando mization and Day planned pSTAT3 (predose [trough] samples only in Phase 2) 0 Treatment laboratory With: assessments pSTAT3 (predose [trough] samples only in Phase 1b) Section 5.2. Delete: Updated to Enrollment/Rando clarify the mization and Day planned laboratory 0 Treatment assessments Section 5.3, Treatment Period/Follow-Up Visits Section 5.2. Replace: Clarified that Enrollment/Rando no need for mization and Day Injection site reaction assessment, predose, and 2 hours post dose predose injection site

| Protocol Date and Ve | ersion: 21 March 2018; V3.0 | |
|---|---|---|
| Section | Description of Changes | Rationale |
| 0 Treatment | With: | reaction assessment at |
| | Injection site reaction assessment, <b>performed at</b> 2 hours postdose | baseline |
| Section 5.3,<br>Treatment<br>Period/Follow-Up<br>Visits | Delete: • Injection site reaction assessments will be performed predose and 2 hours postdose | Clarified that<br>no need for<br>predose<br>injection site<br>reaction<br>assessment at<br>baseline |
| Section 5.3,<br>Treatment | Add: | Updated to |
| Period/Follow-Up<br>Visits | • pSTAT3 (predose [trough] samples only Phase 1b) | clarify the<br>planned<br>laboratory<br>assessments |
| Section 5.4,<br>Safety Follow-Up<br>Visits | | |
| Section 6.6,<br>Pharmacodynamic<br>Assessments | | |
| Section 5.4,<br>Safety Follow-Up<br>Visits | Delete: | Updated to clarify the planned |
| Visits | • pSTAT3 | laboratory<br>assessments |
| Section 6.2.1,<br>Laboratory | Delete: | Updated to clarify the |
| Assessments (Table 3) | Hematology Reticulocytes (%) | planned<br>laboratory |
| | Reticulocytes (70) | assessments |
| Section 6.2.1,<br>Laboratory | Replace: | Updated to clarify the |
| Assessments (Table 3) | Immunogenicity, PD and other Biomarker Tests | planned<br>laboratory |
| (Table 3) | pSTAT3 (predose [trough] samples only, in Phase 2) | assessments |
| | With: | |
| | Immunogenicity, PD and other Biomarker Tests | |
| Section 6.2.1,<br>Laboratory<br>Assessments<br>(Table 3 | pSTAT3 (predose [trough] samples only in Phase <b>1b</b> ) Add: | Text updated<br>to clarify when<br>Coomb's test<br>direct will be |
| | h If clinically indicated for hemolytic anemia. | |
| footnotes) | | collected |

| Section Section | Description of Changes | Rationale |
|---|---|---|
| Section | Description of Changes | Rationale |
| Section 6.2.2.6,<br>Adverse Events of<br>Special Interest | Replace: 2 Injection site reaction, including erythema, pain, and induration With: | Clarify that<br>Grades 2 to 5<br>injection site<br>reactions are<br>AEs of special |
| | 2 Grades 2 to 5 injection site reaction, including erythema, pain, and induration (See APPENDIX 6) | interest |
| Section 6.2.2.6.2,<br>Injection Site<br>Reactions | Replace: | Clarify that<br>Grades 2 to 5 |
| | These may include injection site erythema, pain, and induration. | injection site reactions are |
| | With: | AEs of special interest |
| | These will include Grades 2 to 5 injection site erythema, pain, and induration (see APPENDIX 6). | |
| Section 6.2.7,<br>Injection Site<br>Reaction | Replace: | Clarify that Grades 2 to 5 |
| | Local injection site reactions will be assessed predose and at 2 hours postdose. Injection site reactions should be managed according to the standard of care. Injection site reactions are to be reported as AEs of special interest (see Section 6.2.2.7.3). | injection site<br>reactions are<br>AEs of special<br>interest |
| | With: | |
| | Local injection site reactions will be assessed at 2 hours postdose at baseline, and predose for each injection after baseline. Injection site reactions should be managed according to the standard of care. Injection site reactions, Grades 2 to 5, are to be reported as AEs of special interest (see Section 6.2.2.7.3). | |
| Section 6.3.4.1,<br>SRI-4 Response | Delete: | Differentiate assessment of |
| | Patients will be evaluated for SRI 4 scores at Day 210, with evaluation for sustained reduction of oral CS ( $\leq$ 10 mg/day and $\leq$ Day 0 dose) between Day 120 and Day 210. | SRI-4 and CS usage. |
| Section 6.3.4.1,<br>SRI-4 Response | Delete: | Remove analysis item |
| ord Tresponse | Each patient, after providing their Day 210 visit SRI 4 response, will be evaluated as either a responder or non-responder. | from<br>assessment<br>section |


#### Section **Description of Changes** Rationale Section 6.3.4.2. Delete: Differentiate SRI-5 and SRI-6 assessment of Response The SRI 5 and SRI 6 are evaluated for response at Day 180, along with a SRI-4 and CS sustained reduction of oral CS (≤ 10 mg/day and ≤ Day 0 dose) between usage. Day 120 and Day 210. Remove analysis item from assessment section Section 6.5, Delete: Remove Pharmacokinetic analysis item Assessments PK parameters include the following: from assessment $C_{\text{max}}, T_{\text{max}}, AUC, t_{\downarrow 2}, CL, V_{\text{d}}$ section Plasma concentrations of BOS161721 will be measured using a validated immunoassay. The PK parameters will be calculated from the plasma concentration-nominal time profiles for the IA2 and actual time profiles for the final analysis. The non-compartmental analysis will be performed using appropriately validated PK/PD software. Section 6.6, Delete: Updated to Pharmacodynamic clarify the Assessments planned PD Antibodies: **CC** assessments IgG and IgM and CD4+ count Section 6.8, Delete: Remove Protocol analysis item Deviations Per the statistical analysis plan (SAP), these will be listed by patient and from assessment summarized by deviation category by treatment group. section Section 8, Replace: Updated Statistics (entire section to section) 9 clarify **STATISTICS** statistical analysis plan There are 2 IAs planned for the study. The first IA will be conducted at the time of the POC decision for dose selection. The second IA will be for the study performed for futility (see Section 9.3). Before the first IA, a SAP will be finalized, providing detailed methods for the analyses outlined below. Any deviations from the planned analyses will be described and justified in the final integrated CSR. The following standards will be applied for the analysis unless otherwise specified. Continuous data will be summarized by treatment group using descriptive statistics (number, mean, standard deviation [SD], minimum,

median, and maximum). Categorical data will be summarized by

# Section Description of Changes

Rationale

treatment group using frequency tables (number and percentage).

# 9.1 Sample Size

Sample size in the Phase 1b study is based on operational consideration.

A summary of the power in the trial for the chosen sample size is provided in Table 5, with N=132 randomized 89:43 to the chosen dose for the POC study and placebo, respectively; this includes 12 patients from the MAD study who were in the cohort of the mid or high dose if chosen for the POC study.

Table 5. Sample Size

| Type 1<br>Error<br>(1-<br>Sided) | TRUE<br>Underlying<br>Response Rate<br>(%) | | | Minimum OBSERVED<br>Response Rates<br>Yielding Statistical<br>Significance | |
|---|---|---|---|---|---|
| | Placebo | Treat<br>ment | Overall<br>Power | Placebo | Treatment |
| | 40 | 60 | 0.54 | | |
| 0.025 | 40 | 65 | 0.75 | 40 | 60 |
| | 40 | 70 | 0.9 | | |
| 0.05 | 40 | 60 | 0.63 | | |
| | 40 | 65 | 0.81 | 40 | 58 |
| | 40 | 70 | 0.93 | | |

Total sample size of approximately 156 patients is planned for analysis, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Note that approximately 36 dropouts are assumed.

#### 8.2 Statistical Methods

# 9.2.1 Analysis Populations

The primary efficacy analysis will be based on the full analysis set (FAS), defined to be all patients with at least 1 baseline and post-baseline efficacy evaluation. A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be identified based on blinded data prior to unblinding the final analysis dataset. Safety analyses will be based on all patients who receive test treatment. Pharmacokinetic analysis will be conducted on the PK analysis set (PK), defined as the FAS with sufficient concentration data for the calculation of PK parameters. All analyses will combine data from the MAD and POC studies and focus on the active treatment dose chosen for the POC study versus placebo. The 0.05 1-sided type 1 error level is included for POC, and the 0.025 1-sided type 1 error level for potential use of this trial to support regulatory filing.


# Section Description of Changes

Rationale

#### 9.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized via appropriate summary statistics by treatment group and overall, for each phase of the trial.

#### 9.2.3 Primary Endpoint(s)

The proportion of patients who achieve treatment response (measured by SRI-4 at Day 210 along with a sustained reduction of oral CS) will be analyzed via Cochran-Mantel-Haenszel (CMH) analysis. The primary endpoint will be analyzed on the FAS and if needed the PP analysis set. In addition, missing values will be addressed by employing a last observation carried forward (LOCF) analysis and/or other appropriate analytic approaches as a sensitivity analysis. Details will be available in the SAP.

#### 9.2.4 Secondary Endpoint(s)

Binary efficacy endpoints will be assessed via CMH analysis. Continuous efficacy endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-by-time interaction, baseline covariate, and covariate-by-time interaction. The secondary efficacy endpoint will be analyzed on the FAS and if needed the PP analysis set. Details will be available in the SAP.

#### 9.2.5 Analysis of Safety

#### 9.2.5.1 Safety Analysis

Safety analyses will be performed on the Safety Analysis Set. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. Incidences (number and percent) of AEs will be presented by treatment group. Incidences of AEs will also be presented by maximum severity and relationship to study medication. For the MAD study, the placebo patients from each cohort will be combined for the summaries. If there is a clear increase in AE rates for placebo patients across the cohorts, the AEs will also be summarized by cohort.

AEs will be summarized by counts and percentages of patients by treatment group. Laboratory data and vital signs will be summarized by treatment group as summary statistics for value and change from baseline at each individual time point. Summary statistics will include n, arithmetic mean, median, arithmetic SD, minimum, and maximum.

Additional safety parameters will be analyzed descriptively by treatment group. Descriptive statistics (n, mean, standard deviation (SD), median, minimum, maximum) will be calculated by treatment group and time point for continuous variables. Frequencies and percentages will be presented by treatment group for categorical and ordinal variables.

# Section Description of Changes

Rationale

#### 9.2.5.2 Data Monitoring Committee

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for anti-IL-21 mAb. The recommendations made by the DMC (ie, dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.

The DMC will have access to unblinded treatment information during the clinical trial. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of an anti-IL-21 mAb treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.

- 9.2.6 Pharmacokinetic and Pharmacodynamic Data
- 9.2.6.1 Analysis of Pharmacokinetic Data

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:

- A listing of all plasma BOS161721 concentrations by patient at actual times post dose;
- A descriptive summary of plasma BOS161721 concentrations.
   Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.

Details will be available in the SAP.

9.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Binary PD endpoints will be assessed for the FAS population. Binary PD endpoints will be assessed via CMH analysis. Continuous PD endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-


# Section Description of Changes

Rationale

by-time interaction, baseline covariate, and covariate-by-time interaction. Normality will be assessed via diagnostic residual plots and Shapiro-Wilk statistic, but not as a formal statistical test of normality. If substantial departures from normality are observed, transformation will be used (eg, log and/or rank).

Details will be available in the SAP.

9.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints.

Details will be available in the SAP.

#### 9.3 Interim Analysis and Power

Two IAs are planned for this study. The initial IA will be conducted at the time of the POC decision for dose selection.

The second IA will be performed for futility. IA2 is planned to be conducted at Day 90 when SRI-4 response is determined for approximately 60 patients (including all patients at the same dose level/matching placebo from the MAD study) after completing 3 months of treatment. The purpose of the IA2 is to assess if the trial could stop for an early futility conclusion, or continue. Since there is no plan to stop the trial for an early efficacy conclusion, there is no impact on the type 1 error. If that intention changes, then p < 0.0001 is required for an early efficacy conclusion at the IA2 in order to not impact the planned type 1 error level.

Nominal time profiles will be used for calculating PK parameters in the IA2. Details will be available in the SAP.

With:

#### 8 STATISTICS

The following analyses are planned:

- An IA will be performed during the last cohort of the MAD phase to determine dose selection for the POC phase.
- The final analysis will be performed when all patients have completed the safety follow-up or withdrawn from the study.
- Safety analyses will be performed for DMC reviews throughout the study to evaluate dose escalation decisions and accumulating

Updated to clarify that single alpha for a single primary hypothesis at a significance


## Section Description of Changes

#### Rationale

safety data. The frequency and details of the content and format of the safety review meetings will be described in the SAP and/or DMC charter.

level is acceptable for PoC study.

All statistical analyses will be performed using Statistical Analysis Software (SAS®) Version 9 or higher.

The following standards will be applied for the analysis unless otherwise specified. Data will be summarized descriptively by treatment and overall for each study phase. For the MAD phase, BOS161721 will be summarized overall and by each dose level, and placebo patients from each cohort will be combined. Select parameters will be summarized using patients from both study phases. Statistical testing will be performed on data from the Phase 2 study only.

Continuous data will be summarized using number, mean, standard deviation (SD), 25th and 75th percentiles, minimum, median, and maximum. Categorical data will be summarized by treatment group using frequency tables (number and percentage). Time to event data will be summarized using counts, medians, 25th and 75th percentiles, and standard error. All data will be listed for all patients.

Statistical inference will be based on a 2-tailed test with an overall 0.10 level of significance, unless stated otherwise.

The effects of noncompliance, background therapy use, treatment discontinuations, premature withdrawal from study and covariates will be assessed to determine the impact on the general applicability of results from this study. Exploratory analyses of the data will be conducted as deemed appropriate. Any deviations from the planned analyses will be described and justified in the final integrated CSR.

Protocol deviations and prohibited medications that define medication failures will be fully assigned and documented before database lock and unblinding.

Further details of the analysis, including the handling of missing data, transformations and other data handling procedures will be provided in the SAP.

#### **8.**1 Sample Size

Sample size in the Phase 1b study is based on operational consideration.

The sample size in the Phase 2 study is based on the primary endpoint, SRI-4 Response at Day 210. Approximately 156 additional patients will be randomized in a 2:1 ratio to BOS161721 versus placebo to achieve 132 evaluable subjects in the FAS. This assumes 24 subjects will drop prior to having received treatment and an evaluable post-baseline efficacy measure. Enrollment and randomization will be monitored in a blinded fashion and increased if needed to ensure at least 132 subjects are randomized into the FAS.

Text updated to express in terms of power for selected sample size and primary hypothesis

#### Section

## **Description of Changes**

A total of 132 subjects randomized provides more than 80% power to detect a treatment difference of 25% in SRI-4 response rates at Day 210, based on a targeted 2-sided significance level of 10% and using a 2-sided Pearson's chi-squared test. This assumes of a response rate of 65% for BOS161721 and 40% for placebo, where missing data at Day 210 is carried forward from most recent non-missing result and subjects are treated as a non-responder if a prohibited medication defined as a medication failure occurs.

#### **8.2** Statistical Methods

#### **8.2.1** Analysis Populations

The primary efficacy analysis will be based on the FAS, defined as all patients who receive at least 1 dose of study treatment and have at least 1 evaluable post-baseline efficacy evaluation. FAS analyses will be conducted on the basis of the randomized treatment.

A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be identified based on blinded data prior study to unblinding. PP analyses will be conducted on the basis of the randomized treatment.

Safety analyses will be based on the safety analysis set (SS), defined as all patients who receive at least 1 dose of study treatment. Safety analyses will be conducted on the basis of actual treatment received.

Pharmacokinetic analysis will be conducted on the PK analysis set, defined as the FAS with sufficient concentration data for the calculation of PK parameters.

## **8**.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized **using all** randomized patients.

#### **8**.2.3 Primary **Efficacy** Endpoint(s)

The proportion of patients who achieve a SRI-4 response at Day 210 will be assessed via Pearson's chi-squared analysis. The primary efficacy endpoint will be analyzed using the FAS and if needed repeated in the PP analysis set. Missing values will be addressed by employing a last observation carried forward (LOCF) analysis. Other imputation methods may be employed as a sensitivity analysis and will be described in the SAP. Additional analyses exploring impact of baseline factors such as baseline disease severity, race, and other characteristics may be performed.

Patients that received prohibited medications or unallowable CS usage as described in Section 4.6 will be considered "medication failures" and will be treated as non-responders for the primary

#### Rationale

test, as well as describe alpha, beta, treatment effect assumptions used, and statistical test used for power calculation.

Text updated to clarify that CMH is stratified analysis, and no stratification factors were used at

#### Section

## **Description of Changes**

efficacy analysis. Patients that received an allowable CS burst but having missing data at Day 210 will considered a medication failure and will be treated as non-responders for the primary efficacy analysis. The determination of medication failures will be reviewed using blinded data and finalized prior to unblinding.

The superiority of BOS161721 relative to placebo will be evaluated. If the proportion of SRI-4 responders for the selected POC dose in BOS161721 arm is higher than that of the placebo arm, then BOS161721 will be considered superior to placebo if the 2-sided p-value is less than or equal to 0.10. Secondary and exploratory endpoints for this POC study will be evaluated based on the same statistical hypothesis.

## **8.2.4** Secondary Efficacy Endpoint(s)

Binary efficacy endpoints will be assessed via Pearson's chi-squared analysis. Continuous efficacy endpoints will be assessed via analysis of variance (ANOVA) or analysis of covariance (ANCOVA) and treatment will be compared using the F-test. Repeated measures mixed models may be performed to evaluate data collected at each visit and overall. Time-to-event endpoints will be assessed via Kaplan-Meier methodology and treatment will be compared using the log-rank test. The secondary efficacy endpoints will be analyzed on the FAS and if needed repeated in the PP analysis set. Details including handling of missing data and "medication failures" will be available in the SAP.

#### **8**.2.5 Analysis of Safety

#### 8.2.5.1 Safety Analysis

Safety analyses will be performed on the SS. AE data will be coded to system organ class and preferred term using MedDRA. The number and percentage of patients experiencing any treatment-emergent AE, overall, and by system organ class an preferred term, will be tabulated. Treatment-emergent AEs will also be summarized by severity and relationship.

Concomitant medications will be coded using the WHO Drug dictionary. Observed values and changes from baseline in vital signs, ECG readings, and hematology and clinical chemistry parameters will be summarized at each individual visit.

- **8**.2.6 Pharmacokinetic and Pharmacodynamic Data
- **8**.2.6.1 Analysis of Pharmacokinetic Data

PK parameters will be calculated from concentration data collected during the MAD Phase 1b using non-compartmental analysis and include the following:

#### Rationale

randomization. Population is expected to be relatively homogenous, so Pearson chisquare as primary and secondary analyses may be conducted with factors for adjustment.

Text updated to simplify and maintain consistency with binary endpoints. Allows more flexibility in handling missing data.

# Section Description of Changes

Rationale

•  $C_{max}$ ,  $T_{max}$ , AUC,  $t_{\frac{1}{2}}$ , CL,  $V_d$ 

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:

- A listing of all plasma BOS161721 concentrations by patient at actual times post dose;
- A descriptive summary of plasma BOS161721 concentrations.
   Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.

#### **8**.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Exploratory analyses examining the relationship between PD parameters and PK concentration and PK parameters will be performed.

8.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints

## **8.3** Interim Analysis and Power

One IA is planned for this study and will be conducted at the time of the POC decision for dose selection.

Since there is no **IA during the POC phase**, there is no impact on the type 1 error.

The futility analysis was removed due to the modest size of the trial but more importantly because the least reliable data (high placebo response) is known to occur during the first half of

#### Section

## **Description of Changes**

#### Rationale

the study (before week 24) when futility analysis was planned

# Section 9.2, DMC Replace:

Clarification and to remove redundant text

The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) suggest dose for POC portion of the study.

The DMC considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

#### With:

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for BOS161721. The recommendations made by the DMC (ie, dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.

The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) suggest dose for POC portion of the study as described in Section 3.1.1.3.

The DMC considers study-specific data as well as relevant background

# Section Description of Changes

Rationale

knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

The DMC will have access to unblinded treatment information during the clinical trial. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of BOS161721 treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.
#### Section

#### **Description of Changes**

#### Rationale

#### Appendix 1, Names of Study Personnel

Replace:



Updated to represent change in personnel

#### With:



#### Appendix 4, Medication Washout Periods

Replace:

| Medication | Discontinuing Prior to Signing<br>Consent |
|------------|-------------------------------------------|
| Belimumab | 48 weeks |

Updated text to clarify when medication had to be discontinued prior to study initiation

#### With:

| Medication | Discontinuing Prior to Signing<br>Consent |
|------------|-------------------------------------------|
| Belimumab | 24 weeks |

Appendix 5, BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA) Replace:





Section Description of Changes Rationale



Section Description of Changes Rationale



Appendix 6, INJECTION SITE REACTION GRADING SCALE Add:

| Adverse event<br>Injection site<br>reaction | Grade 1 | Grade 2 | Grade 3 | Grade<br>4 | Grade<br>5 |
|---|---|---|---|---|---|
| Definition: A disorder characterized by an intense adverse reaction (usually immunologic) developing at the site of an injection | Tenderness with or without associated symptoms (eg, warmth, erythema, itching) | Pain;<br>Lipodystr<br>ophy;<br>Edema;<br>phlebitis | Ulceratio<br>n or<br>necrosis;<br>Severe<br>tissue<br>damage;<br>Operativ<br>e<br>intervent<br>ion<br>indicated | Life-<br>threat<br>ening<br>conseq<br>uences<br>;<br>urgent<br>interve<br>ntion<br>indicat<br>ed | Death |
| Pain | Mild pain | Moderat<br>e pain;<br>limiting<br>instrume<br>ntal ADL | Severe<br>pain;<br>limiting<br>self-care<br>ADL | - | - |
| Rash<br>maculopapular/ | Macules/pa<br>pules | Macules/<br>papules | Macules/<br>papules | - | - |

Added table to clarify the grading scale for injection site reactions

#### Section Description of Changes Rationale

| Erythema/Indur ation | covering<br><10% BSA | covering<br>10% - | covering > 30% | |
|---|---|---|---|---|
| ation | with or | 30% BSA | BSA with | |
| 5 | without | with or | or | |
| Definition: A | symptoms | without | without | |
| disorder | | | associate | |
| characterized by | (eg, | symptom | d | |
| the presence of | pruritus, | s (eg, | ~ | |
| macules (flat) | burning, | pruritus, | symptom | |
| and papules | tightness) | burning, | s; | |
| (elevated). Also | Erythema | tightness | limiting | |
| known as | covering | ); limiting | self-care | |
| morbillform | <10% BSA | instrume | ADL | |
| rash, it is one of | with or | ntal ADL; | | |
| the most | without | Erythema | Erythema | |
| common | symptoms | 30% BSA | covering | |
| cutaneous | (eg, | with or | > 30% | |
| adverse events, | pruritus, | without | BSA with | |
| frequently | burning, | symptom | or | |
| affecting the | tightness) | s (eg, | without | |
| upper trunk, | | pruritus, | associate | |
| spreading | | burning, | d | |
| centripetally, | | tightness | symptom | |
| and associated | | ); limiting | s; | |
| with pruritus. | | instrume | limiting | |
| | | ntal ADL | self-care | |
| | | | ADL | |
| | | | | l |

ADL = active daily living



# A RANDOMIZED DOUBLE-BLIND PHASE 1b/2 COMBINED STAGGERED MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF LIMITED STANDARD OF CARE

**SPONSOR** Boston Pharmaceuticals, Inc.

55 Cambridge Parkway, Suite 401

Cambridge, MA 02142

United States of America (USA)

INVESTIGATIONAL COMPOUND: BOS161721

PROTOCOL NUMBER: BOS161721-02

PHASE Phase 1b/2

INVESTIGATIONAL NEW DRUG (IND)

**NUMBER:** 

131796

ORIGINAL PROTOCOL DATE: 05 October 2017

**VERSION NUMBER:** V2.0 (Amendment 1)

**VERSION DATE:** 08 November 2017

BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02

#### CLINICAL PROTOCOL APPROVAL FORM

Protocol Title: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

Study No: BOS161721-02

Original Protocol Date: 05 October 2017 Protocol Version No: v2.0 (Amendment 1) Protocol Version Date: 08 November 2017

This study protocol was subject to critical review and has been approved by sponsor. The information contained in this protocol is consistent with:

- The current risk-benefit evaluation of the investigational product.
- The moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (APPENDIX 2), and principles of Good Clinical Practices (GCP) as described in 21 Code of Federal Regulations (CFR) parts 50, 54, 56 and 312 and according to applicable local requirements.

The investigator will be supplied with details of any significant or new findings, including adverse events, relating to treatment with the investigational product.

I agree with these statements and indicate my approval by signature for this protocol:

| Name and Title | Signature | Date |
|---|---|---|
| PPD, MD Vice President, Clinical Development Boston Pharmaceuticals | PPD | |
| PPD Clinical Operations Lead Boston Pharmaceuticals | PPD | |
| PPD , MD, PhD Vice President, Clinical Development and Safety Officer Boston Pharmaceuticals | PPD | |

## **SUMMARY OF CHANGES**

| Section | <b>Description of Changes</b> | Rationale |
|---|---|---|
| Global | Change: | Administrative |
| | Changed Version number from V1.0 to <b>V2.0 (Amendment 1)</b> and Version date from 05 October 2017 to <b>08 November 2017</b> . | |
| Global | Change: | For clarity, site visits are based on study day |
| | Removed use of "Months" and "Weeks" to describe study site visits and dosing. Changed to <b>Day X</b> throughout protocol. | number only. |
| Global | Change: | Clarification (as dose is given every 30 days) |
| | Changed randomization day from Day 1 to <b>Day 0</b> . | given every 30 days) |
| Global | Made administrative and editorial (formatting, typographical, and grammatical) updates. | Administrative |
| PROTOCOL | Replace: | Clarification and updated with new safety data. |
| SUMMARY, Background and Rationale Section 1.2.2.3, Clinical Studies | Overall, there were no clinically significant findings from this study; there were no serious adverse events (SAEs), deaths, or discontinuations due to AEs during the study, AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. | |
| | With: | |
| | Overall, there were no clinically significant findings from this study, following an interim cut and review of the data at Day 90 postdose. Adverse events reported as related to the study drug, particularly infections, were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. There was 1 serious adverse event (SAE; death due to pulmonary embolism) that occurred 127 days after a single administration of 240 mg SC dose of BOS161721. The causality of this single SAE was not attributed to study drug and further information can be found in the Investigator's Brochure. | |


#### Section **Description of Changes** Rationale **PROTOCOL** Delete: Clarification to correct SUMMARY, level of exposure Study Design Each of the 3 doses (20 mg, 60 mg, and 120 mg) selected for the MAD study are projected not to exceed the mean peak levels or Section 1.2.3, exposures of that achieved in the SAD study following the single Study Dose Section 240 mg SC dose. Section 4.1.1, Multiple Ascending Dose Phase 1b Study **PROTOCOL** Replace: Removed erroneous SUMMARY, text and added clarity Study Design Similarly, after 8 of the 12 patients in Cohort 2 have received that Boston 2 doses and have completed 2 weeks of follow-up after the Pharmaceuticals will review data along with second dose, Cohort 3 begins dosing (based on the dose level determined after DMC evaluation of the safety and tolerability DMC for POC Dose data from Cohort 2 and Cohort 1). Two weeks after the last selection. patient in Cohort 3 receives the second dose, the DMC will conduct a data review for the first interim analysis (IA1) to determine which dose will be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available when the last patient in Cohort 3 reaches 60 days (dose 2). This dose will not exceed doses tested during the MAD study. With:

Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after DMC evaluation of the safety and tolerability data from Cohort 2 and Cohort 1. Two weeks after the last patient in Cohort 3 receives the second dose, the DMC and Boston Pharmaceuticals will conduct a data review for the first interim analysis (IA1). At that time, a decision will be made to suggest which dose should be carried forward into the POC Phase 2 study. This dose will not exceed doses tested during the MAD study.

Confidential

| Section | Description of Changes | Rationale |
|---|---|---|
| PROTOCOL<br>SUMMARY, | Add: | Clarification to allow flexibility in exact |
| Study Design | approximately 156 patients | number enrolled. |
| Section 4.1.2.2,<br>POC Study Design | | |
| Section 9.1, Sample Size | | |
| PROTOCOL<br>SUMMARY, | Replace: | Second period for allowed CS "burst" |
| Study Design | One oral CS "burst" for increased SLE disease activity may occur during the study either between Weeks 1 and 8 or between Weeks 16 and 20. | removed as it conflicts with study endpoints. |
| | With: | |
| | One oral CS "burst" for increased SLE disease activity may occur during the study between <b>Day 0</b> and <b>Day 60</b> . | |
| PROTOCOL<br>SUMMARY, | Replace: | Replaced weeks with days to be consistent |
| Study Design | Tapering may occur after randomization except within 8 weeks of the primary (Week 28) and secondary (Week 16) endpoint | with protocol. |
| Section 5.6.1, Oral<br>Corticosteroid | assessments. | |
| Dose | With: | |
| | Tapering may occur after randomization except within <b>60 days</b> of the primary ( <b>Day 210</b> ) and secondary ( <b>Day 120</b> ) endpoint assessments. | |
| Section 1.2.3;<br>Study Dose Section | Replace: | Clarification that Boston Pharmaceuticals |
| Study Dose Section | In addition, the DMC will conduct a data review for the first interim analysis (IA1) to determine which dose will be carried forward into the proof of concept (POC) Phase 2 study. | will review data along with DMC for POC Dose selection. |
| | With: | |
| | In addition, the DMC and Boston Pharmaceuticals will conduct a data review for the first interim analysis (IA1). At that time, a decision will be made to suggest which dose should be carried forward into the proof of concept (POC) Phase 2 study. | |

#### Section

#### **Description of Changes**

#### Section 1.2.4, Risk-Benefit Assessment

#### Replace:

Two weeks after the last patient in Cohort 3 receives the second dose, the DMC will conduct a data review for the IA1 to determine which dose will be carried forward into the POC Phase 2 study.

#### With:

Two weeks after the last patient in Cohort 3 receives the second dose, the DMC and Boston Pharmaceuticals will conduct a data review for the IA1. At that time, a decision will be made to suggest which dose should be carried forward into the POC Phase 2 study.

#### Section 4.1.1.1; Dose Escalation for the MAD Study

#### Delete:

Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing (based on the dose level determined after DMC evaluation of the safety and tolerability data from Cohorts 1 and 2). Two weeks after the last patient in Cohort 3 receives the second dose, the DMC will conduct a data review for the IA1 to determine which dose will be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available when the last patient in Cohort 3 reaches 60 days (dose 2).

#### Section 4.1.1.1; Dose Escalation for the MAD Study

Replace:

If > 3 patients discontinue the study in a cohort, he/she will be replaced.

With:

If > 3 patients discontinue the study in a cohort, he/she **may** be replaced.

# Section 4.1.1.2;

Dose Limiting Toxicity (DLT)

#### Delete:

Investigators should always manage their patients according to their medical judgment which may include interruption of study drug based on the particular clinical circumstances.—All dose modifications/adjustments must be clearly documented in the patient's source notes and electronic Case Report Form (eCRF).

#### Rationale

Clarification that Boston Pharmaceuticals will review data along with DMC for POC Dose selection.

Removed, as this information does not fit this section.

Clarified statement as it is not definitive that these patients would be replaced.

Dose modifications/ adjustments are not allowed in this study.

#### Section

#### **Description of Changes**

#### Section 4.1.1.3:

**DMC** 

Recommendations

#### Replace:

For the POC study, the DMC will conduct a data review for the IA1 to determine which dose will be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available when the last patient in Cohort 3 reaches 60 days (dose 2). Details are provided in the DMC Charter.

#### With:

For the POC study, the DMC and Boston Pharmaceuticals will conduct a data review for the IA1 to suggest which dose should be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available at the time the last patient in Cohort 3 completes the Day 44 visit (2 weeks after dose 2). Details are provided in the DMC Charter.

#### Section 4.1.2.1; BOS161721 Dose

#### Replace:

The optimal dose evaluation is chosen based on MAD Phase 1b safety results. The dose will be communicated by a letter to site investigators participating in the POC Phase 2 study, and to the IRB/IEC. Once the POC dose decision has been made, screening for the POC study can begin.

#### With:

The optimal dose evaluation is chosen based on MAD Phase 1b safety, tolerability, immunogenicity, and PK and PD data. The dose will be communicated by a letter to site investigators participating in the POC Phase 2 study, and to the IRB/IEC.

#### Section 4.2, Study Schematic, Figure 2

#### Change:

Study schematic was updated to reflect use of "Days" for dosing as well as a correction to the time point for dose escalation (change from "Day 60" to "Day 44").

#### Rationale

Corrected error, data cut for the DMC review will be 2 weeks after dose 2 (Day 44 visit).

Updated for consistency with rest of protocol.

To reflect changes made to protocol body.

| Section | Description of Changes | Rationale |
|---|---|---|
| Section 4.3,<br>Schedule of | Change: | Reorganized for better clarity |
| Assessments,<br>Table 1, Table 2 | Schedule of Assessments was reorganized so that all assessments are categorized as: General, Safety, Efficacy, Laboratory, or PK Labs. Footnotes were relettered accordingly. | |
| Section 4.3,<br>Schedule of<br>Assessments,<br>Table 2 | Change: Removed columns for Day 7 and Day 44 in POC Schedule of Assessments. | These visits are not applicable in the POC portion of this study. |
| Section 4.3,<br>Schedule of | Change: | Safety information should be collected |
| Assessments,<br>Table 1, Table 2 | Added assessments on Days 7 (MAD only), 187, and 195 for concomitant medications, AEs and SAEs, and injection site reactions. | even on PK-only visits. |
| Section 4.3,<br>Schedule of | Delete: | Estradiol is removed as FSH is sufficient to |
| Assessments, Table 1, Table 2 | FSH and estradiol (postmenopausal women) | determine menopause |
| Section 6.1,<br>Screening | | |
| Section 7.2.1,<br>Laboratory<br>Assessments,<br>Table 3 | | |
| Section 4.3,<br>Schedule of | Add: | Clarification |
| Assessments, Table 1, Table 2, footnote g | Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, | |
| Section 7.2.3, Vital Signs | 187, and 195). | |
| Section 4.3,<br>Schedule of | Replace: | Clarification |
| Assessments,<br>Table 1, Table 2,<br>footnote h | Clinical laboratory assessments will include a fasting glucose and lipid panel during screening and Week 28. | |
| <del></del> | With: | |
| | Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting. | |

Rationale

BOS161721 Clinical Study Protocol: BOS161721-02

| Section | Description | ~ 4 |
|---------|-------------|-----|

#### Section

#### **Description of Changes**

#### Section 5.6.1, Oral Corticosteroid

Dose

Delete:

A maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed during the study either between Day 0 and Day 60 or between Weeks 16 and 20, according to the following:

Second period for allowed CS "burst" removed as it conflicts with study endpoints.

Section 5.6.1, Oral Corticosteroid Dose

Delete:

- An oral CS "burst" between Week 16 and Week 20 (an increase of ≤ 20 mg/day prednisone or equivalent), which must be tapered down to a maximum of 10 mg/day within 2 weeks of initiation of the "burst".
  - Alternatively, a single IM dose of methylprednisolone (40 mg or equivalent) is permitted.

Second period for allowed CS "burst" removed as it conflicts with study endpoints.

Section 5.6.2, Other Prohibited and/or Restricted

Treatments

Replace:

Prohibited and/or restricted medications taken prior to study drug administration in the study are described below, and washout requirements are provided in APPENDIX 4.

Clarification – this list includes not only prohibited medication prior to first dose, but also restrictions during the study.

With:

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in APPENDIX 4.

Section 5.8.2, Exception for Non-Responders

Delete:

#### 5.8.2 **Exception for Non-Responders**

Patients will be classified as non-responders if they (1) receive a second rescue medication at any time in the study or (2) take rescue medications between Week 8 and Week 16 or between Week 20 and Week 28 (as described in Section 5.6.1). If a patient has been deemed a non responder, they will discontinue from treatment and all End of Treatment assessments will be performed. The patient will then enter the safety follow-up period. The use of rescue medications in the case of non responders is not to be considered a protocol violation (exclusion criteria 8). Protocol violations will be identified based on blinded data prior to unblinding the final analysis dataset.

Section deleted. Patients requiring corticosteroid outside of the protocol allowed time should be included in safety analysis and therefore continue in study. Use of corticosteroid excluded from protocol windows would be documented as protocol violations.

Section 6.1, Screening

Delete:

Screening will be the same for both the MAD and POC studies. Screening for the POC study cannot begin until the POC dose decision has been made.

Screening for POC study can begin while dose decision is being made.

| Section | Description of Changes | Rationale |
|---|---|---|
| Section 6.1,<br>Screening | Add: • Chest x-ray | Chest x-ray was added as it was missing from V1.0 list of |
| | <ul> <li>Laboratory evaluations (nonfasting):</li> </ul> | assessments. "(nonfasting)" was added as clarification. |
| Section 6.2,<br>Enrollment/Rando<br>mization and Day 0<br>Treatment | Add: • Laboratory evaluations (fasting): | Clarification |
| Section 6.3,<br>Treatment<br>Period/Follow-Up<br>Visits | Replace: See Section 4.3 for allowable windows for each visit. The following procedures will be performed at every study drug administration visit (Weeks 4, 8, 12, 16, 20, and 24) and follow-up visits during the treatment period (Weeks 2 and 6): With: The following procedures will be performed as indicated in the Schedule of Assessments (Table 1 and Table 2). See Schedule of Assessment tables for allowable windows for each visit. | Clarification |
| Section 6.3, Treatment Period/Follow-Up Visits Section 6.3, Treatment Period/Follow-Up | Change: Based on change above (ie, cross-reference to Schedule of Assessments), removed timing of assessments from bulleted listed. Replace: Hematology and chemistry assessments will be performed at | Clarification Clarification |
| Visits | <ul> <li>Weeks 4 and 6 (Visits 4 and 5) for the MAD study, only, and at Weeks 8, 12, 16, 20, and 24 (Visits 6 through 10) for both studies.</li> <li>With:</li> <li>Fasting hematology and chemistry assessments</li> </ul> | |
| Section 6.4, Safety<br>Follow-Up Visits | Add: These visits will include the following assessments as indicated in the Schedule of Assessments (Table 1 and Table 2): | Clarification |
| Section 6.4, Safety<br>Follow-Up Visits | Change: Based on change above (ie, cross-reference to Schedule of Assessments), removed timing of assessments from bulleted listed. | Clarification |

## Section Section 6.4, Safety Add: Follow-Up Visits Section 7.2.1, Delete: Laboratory

#### **Description of Changes**

Fasting clinical laboratory assessments (hematology and clinical chemistry)

# Assessments

Laboratory/analyte results that could unblind the study (ie, biomarker results) will not be reported to investigative sites or other blinded personnel until the study has been unblinded. Urinalysis will be performed on midstream, clean catch

specimens.

Section 7.2.1, Laboratory Assessments

Add:

Endpoint analyses will be based on changes from baseline assessments at Days 120 and 210.

Section 7.2.1, Laboratory Assessments, Table 3

Add:



Section 7.2.1.1. Pregnancy testing Replace:

Urine pregnancy tests will also be routinely repeated at study drug administration visits (Visits 2, 4, 6, 7, 8, 9, and 10) prior to study drug administration, and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be withdrawn from study drug but may remain in the study for safety monitoring.

With:

Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 6.4).

#### Rationale

Clarification

Text removed as

**Boston Pharmaceuticals** will be reviewing biomarker data for POC dose selection.

Moved from redundant laboratory assessment section that was deleted from protocol.

Clarification (genotype needed to establish gene signature)

To clarify how the patient should complete the study. Also removed Visit numbers as beginning of section cross-references Schedule of Assessments.

| Section | <b>Description of Changes</b> | Rationale |
|---|---|---|
| Section 7.2.4,<br>12-Lead<br>Electrocardiograms | Replace: | Clarification |
| | ECG will be performed at screening, and Visits 2, 4, and 7, and 13. | |
| | With: | |
| | ECG will be assessed as specified in the Schedule of Assessments (Section 4.3). | |
| Section 7.2.5, | Replace: | Clarification |
| Physical<br>Examination | The targeted (limited) physical examination will be completed at Visits 3 through 13. | |
| | With: | |
| | The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Section 4.3). | |
| Section 7.2.6,<br>C-SSRS | Replace: | Clarification |
| C-55K5 | The C-SSRS evaluation will be performed at screening, Visit 2 (Day 1) and at Visits 7 and 10 (Weeks 12 and 24, respectively). | |
| | With: | |
| | The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Section 4.3). | |
| Section 7.2.7,<br>Injection Site | Replace: | Clarification |
| Reactions | Patients will be monitored for local injection site reactions at dosing administration visits, Visits 2 (Day 1), Visit 4 (Week 4), and Visits 6 through 10 (Weeks 8, 12, 16, 20, and 24). Patients will also be monitored for local injection site reactions at the safety follow-up visits, Visits 11, 12, and 13 (Weeks 28, 32, and 36, respectively). | |
| | With: | |
| | Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (Section 4.3). | |

| Section | Description of Changes | Rationale |
|---|---|---|
| Section 7.2.8,<br>Immunogenicity | Replace: | Clarification |
| | The serum samples to measure the presence of ADA will be collected as Visits 2, 3, 4, 6, 7, 10, and 13 (Week 0, 2, 4, 8, 12, 24, and 36, respectively). | |
| | With: | |
| | The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (Section 4.3). | |
| Section 7.3,<br>Efficacy | Add: | Clarification (allows for deletion of visit |
| Assessments | All efficacy assessments will be performed at times defined in the Schedule of Assessments (Section 4.3). | days from each subsection). |
| Section 7.3.1,<br>SLEDAI-2K | Delete: | Removed based on cross-reference to |
| SLEDAI-2K | The SLEDAI 2K is completed at screening, at Visit 2, Visit 4, and Visits 6 through 13. | Schedule of Assessments provided in Section 7.3. |
| Section 7.3.2,<br>BILAG 2004 | Delete: | Removed based on cross-reference to |
| BILAU 2004 | The BILAG 2004 is completed at screening, Visit 2, 4, and 6 through 13. | Schedule of Assessments provided in Section 7.3. |
| Section 7.3.3, PGA of Disease Activity | Delete: | Removed based on cross-reference to |
| of Disease Activity | The PGA is completed at screening, Visit 2, 4, and Visits 6 through 13. | Schedule of Assessments provided in Section 7.3. |
| Section 7.3.6,<br>ACR-28 Joint<br>Count | Delete: | Removed based on cross-reference to |
| | The ACR 28 joint count will be performed at screening, Visit 2, 4, and 6 through 13. | Schedule of Assessments provided in Section 7.3. |

#### Section

#### **Description of Changes**

#### Rationale

Section 7.3.7, Laboratory Assessments Delete:

7.3.7 Laboratory Assessments

Deletion of redundant information already presented in Section 7.2.1.

Patients will be evaluated for laboratory parameters as specified in the Schedule of Assessments (Section 4.3), including: Fasting glucose and lipid panels, pSTAT3 (predose samples in Phase 2), total IgG & IgM, complement: CCI , Plasma CCI & & , whole blood for leukocyte immunophenotype and RNA, CCI , and antibodies: (CCI)

Endpoint analyses will be based on changes from baseline assessments at Week 16 and Week 28.

Section 7.4.2, PROs

Add:

Clarification

The PROs include the CCI and will be assessed as specified in the Schedule of Assessments (Section 4.3).

Delete:

The CClassic is completed by patients at screening and Day 1 (Visit 2), Week 4 (Visit 4), Week 8 (Visit 6) through Week 36 (Visit 13).

Delete:

The CCI -is administered at screening, and Day 1 (Visit 2) Week 4 (Visit 4), Week 8 (Visit 6) through Week 36 (Visit 13).

Section 7.5, Pharmacokinetic Assessments Delete:

This language is not applicable under PK section.

PK parameters include the following:

•  $C_{max}$ ,  $T_{max}$ , AUC,  $t_{1/2}$ , CL,  $V_d$ 

In addition to samples collected at the scheduled times, an additional blood sample should be collected from patients experiencing unexpected AEs and/or SAEs and the date and time documented in the cCRF.

Section 7.6, Pharmacodynamic Assessments Add:

Clarification

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (Section 4.3) for each of the following parameters:

| Section | <b>Description of Changes</b> | Rationale |
|---|---|---|
| Section 7.6,<br>Pharmacodynamic<br>Assessments | Change: | Clarification |
| | Based on change above (ie, cross-reference to Schedule of Assessments), removed timing of assessments from bulleted listed. | |
| Section 8.5,<br>Prohibited | Add: | Clarification |
| Concomitant<br>Therapy | Prohibited concomitant medications are discussed in Section 5.6 and APPENDIX 4 and will be listed as protocol violations if taken when not permitted. | |
| Section 9.2.5.2, | Delete: | Removed text, exact details will be provided |
| Data Monitoring<br>Committee | The DMC will have access to unblinded treatment information during the clinical trial.—To prevent inadvertent unblinding of sponsor staff, reports to the DMC will describe each treatment group by a coded identifier rather than actual treatment group assignment. Details regarding management and process of this committee are found in the DMC Charter. | in charter. |
| Section 9.3, Interim<br>Analysis and Power | Delete: | Removed as efficacy data will be reviewed |
| Analysis and Power | Two IAs are planned for this study. The initial IA will be conducted at the time of the POC decision for dose selection. The DMC will review safety and tolerability, and PK/PD/biomarkers for dose selection. Efficacy data will not be reviewed for dose selection so there should be no impact on the type 1 error. | by Boston Pharmaceuticals in order to make informed dose selection decision. |
| Section 9.3, Interim<br>Analysis and Power | Add: | Clarification |
| | Nominal time profiles will be used for calculating PK parameters in the IA2. <b>Details will be available in the SAP.</b> | |
| Section 10.2, DMC | Replace: | Clarification |
| | The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) make a dose recommendation for POC portion of the study. | |
| | With: | |
| | The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) <b>suggest</b> dose for POC portion of the study. | |

# Section 10.4, Informed Consent Replace: Before each patient is enrolled in the clinical study, written informed consent will be obtained from the patient according to the regulatory and legal requirements of the participating country. With: Before each patient undergoes any protocol required assessments or procedure, the written informed consent will be obtained according to the regulatory and legal requirements of the participating country.

#### BOS161721-02

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

#### CONFIDENTIALITY AND INVESTIGATOR STATEMENT

The information contained in this protocol and all other information relevant to BOS161721 are the confidential and proprietary information of Boston Pharmaceuticals, Inc., and except as may be required by federal, state, or local laws or regulation, may not be disclosed to others without prior written permission of Boston Pharmaceuticals, Inc.

I have read the protocol, including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described. I will conduct this study as outlined herein, in accordance with the regulations stated in the Federal Code of Regulations for Good Clinical Practices and International Council for Harmonisation (ICH) guidelines, and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and any amendments, and access to all information provided by Boston Pharmaceuticals, Inc., or specified designees. I will discuss the material with them to ensure that they are fully informed about BOS161721 and the study.

| Principal Investigator Name (printed) | | Signature |
|---------------------------------------|-------------|-----------|
| <br>Date | Site Number | |


BOS161721

Clinical Study Protocol: BOS161721-02

#### PROTOCOL SUMMARY

Title:

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

Indication

Adults with moderately to severely active SLE

Background and Rationale

SLE is a chronic systemic autoimmune disease with considerable heterogeneity in clinical manifestations and disease course. There is evidence that B- and T-cells are critical to the development of the disease, and that T-cell-derived cytokines such as interleukin-21 (IL-21) are involved in the SLE-associated inflammatory pathological response.

BOS161721 is a humanized immunoglobulin G1 (IgG1) triple mutation monoclonal antibody (mAb) intended to have an extended terminal elimination half-life ( $t_{1/2}$ ) that selectively binds to and neutralizes IL-21, which acts on multiple cell types that drive inflammation and autoimmunity. In vivo, BOS161721 inhibits T-cell dependent antigen responses of B-cells and is being developed as a potential treatment for adults with moderately to severely active SLE.

Nonclinical studies have evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), pharmacokinetics (PK), and immunogenicity of BOS161721 administered intravenously (IV) and subcutaneously (SC). The no observed adverse effect levels (NOAELs) in Cynomolgus monkeys were determined to be 100 mg/kg IV and 50 mg/kg SC, the highest doses tested. No SC animals had injection reactions.

In a Phase 1 single ascending dose (SAD) study, BOS161721 was administered IV and SC to healthy male and female adult subjects. This double-blind, placebo-controlled study evaluated 8 ascending dose levels (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) for safety, tolerability, PK, PD and immunogenicity. Overall, there were no clinically significant safety or tolerability findings from this study, following an interim cut and review of the data at Day 90 postdose.

Results from the Phase 1 SAD study informed the dose regimens used for the multiple ascending doses (MAD) Phase 1b study in this trial. The MAD study will involve 3 cohorts. The Phase 2 portion will be a proof of concept (POC) study, where dose selection will be based on the sponsor's assessment of safety, tolerability,

immunogenicity, and PK and PD data from the MAD study of 30 patients treated with BOS161721/placebo. The purpose of the study is to establish safe and effective dosages for adult patients with moderately to severely active SLE.

#### **Objectives:**

#### **MAD Phase 1b Study**

#### **Primary Objective:**

To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20 mg, 60 mg, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose.

#### **POC Phase 2 Study**

#### **Primary Objective:**

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on the SLE Responder Index 4 (SRI-4), with sustained reduction of oral corticosteroids (CS), in adult patients with moderately to severely active SLE on limited background standard of care treatment.

#### **Secondary Objectives:**

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment, including:

- Changes in SLE-specific autoantibody titers
- Changes in complement 3 and 4 (C3 and C4) levels
- Responses on SRI-4, SLE Responder Index 5 and 6 (SRI-5, and SRI-6), with sustained reduction of oral CS
- Response on the British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (BICLA)
- Response on the Cutaneous Lupus Erythematosus Area and Severity Index (CLASI)
- Changes in the SLE Disease Activity Index 2000 (SLEDAI-2K)
- Changes in the American College of Rheumatology (ACR)-28 joint count

#### **Endpoints:**

#### **Phase 1b MAD Study**

#### **Primary Endpoints:**

Evaluation of safety, tolerability, and immunogenicity at each dose level, to determine the optimal dose, will include the recording of the following parameters:

- Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)
- 12-lead electrocardiograms (ECGs)
- Vital signs (blood pressure [BP], heart rate, and temperature)
- Clinical laboratory assessments
- Physical examinations
- Evaluation for anti-drug antibodies (ADAs)

#### **Exploratory Endpoints:**



**Other Endpoints:** 



#### **PRO Endpoints:**



#### **Phase 2 POC Study**

#### **Primary Efficacy Endpoint:**

The primary efficacy endpoint is the proportion of patients who achieve treatment response as measured by the SRI-4 at Day 210, along with a sustained reduction of oral CS ( $\leq$  10 mg/day and  $\leq$  Day 0 dose) between Day 120 and Day 210.

#### **Secondary Efficacy Endpoints:**

- The proportion of patients who achieve treatment response for the SRI-5 and SRI-6 at Day 210, along with a sustained reduction of oral CS (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210
- Changes from baseline in dsDNA, ANA, SSA, SSB, RNP, Sm, APL autoantibodies, at Day 120 and Day 210
- Changes from baseline in C3 and C4 levels at Day 120 and Day 210
- Changes from baseline in the SLEDAI-2K at Day 210
- Time to BILAG A or B flare
- Changes from baseline in the CLASI at Day 210
- The proportion of patients with a BICLA response at Day 210
- The proportion of patients with CLASI response at Day 210

- Changes from baseline (percentage) in swollen joints and tender joints ACR-28 joint count
- Assessment of safety, tolerability, and immunogenicity as described for the primary endpoint in the MAD Phase 1b study

#### **Exploratory Endpoints:**

• CCI

#### **Other Endpoints:**

- CCI
- CCI
- CCI

#### **PRO Endpoints:**

- CCI
- CCI

#### **Study Design:**

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of multiple SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly. The trial will consist of a staggered MAD Phase 1b and POC Phase 2 studies. Both studies will be double-blinded with each patient having the same number of doses (7), and visits; the duration will be 180 days, followed by a 90-day follow-up safety observation period.

The MAD Phase 1b study phase will consist of 3 cohorts, with Cohort 1 containing 6 patients, where 5 of these patients will receive BOS161721 (active), and 1 will receive placebo. Cohorts 2 and 3 will each contain 12 patients, including 9 active and 3 placebo

patients. Dose selection for each cohort is based on 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. Each of the 3 doses (20 mg, 60 mg, and 120 mg) selected for the MAD study are projected not to exceed the mean exposure of that achieved in the SAD study following the single 240 mg SC dose. Each patient may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180.

The MAD study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after a data monitoring committee [DMC] evaluates the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after DMC evaluation of the safety and tolerability data from Cohort 2 and Cohort 1. Two weeks after the last patient in Cohort 3 receives the second dose, the DMC and Boston Pharmaceuticals will conduct a data review for the first interim analysis (IA1). At that time, a decision will be made to suggest which dose should be carried forward into the POC Phase 2 study. This dose will not exceed doses tested during the MAD study.

For the POC study, approximately 156 patients will be randomized to active or placebo groups in a 2:1 ratio. As in the MAD study, each patient in the POC study may receive a total of 7 SC monthly doses on Days 0, 30, 60, 90, 120, 150, and 180. A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). One oral CS "burst" for increased SLE disease activity may occur during the study between Day 0 and Day 60. Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits. Tapering may occur after randomization except within 60 days of the primary (Day 210) and secondary (Day 120) endpoint assessments. Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant otherwise the patient will be declared a non-responder in efficacy assessments.

Data from 60 patients, including the 12 from the MAD study, or 6 fewer if the low dose is chosen, who are in the cohort of the chosen dose for the POC study who complete 3 months of treatment will be used in a second IA (IA2) at Day 90 to assess if the trial could stop for an early futility conclusion. If futility is not claimed in the IA2, the POC study will continue to approximately 156 patients.

Following the 6-month treatment period, primary and secondary efficacy endpoints will be assessed for each patient, after providing their Day 180 disease activity assessments. DMC monitoring will be conducted periodically throughout the study as described in the DMC charter.

# Main Criteria for Inclusion and Exclusion

#### **Inclusion Criteria:**

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion OR Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Sm above the normal level as determined by the central laboratory
  - c. C3 or C4 below normal as determined by the central lab
- 5. At screening, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at

least 1 of the following clinical components:

- a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
  - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia and leukopenia
  - ii. Points from lupus headache and organic brain syndrome are also excluded
- 7. Patients must have at least 1 of the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 5.4
  - c. If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores
- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization)
- 9. Women of childbearing potential (WOCBP; see Section 5.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening.

Urine pregnancy test must be negative prior to first dose

- b. Must not be breastfeeding
- c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS1617219 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

#### **Exclusion Criteria**

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment

- with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count  $< 500/\mu$ L at screening
- 16. Platelets  $< 50,000/\text{mm}^3$  (50  $\times$  10<sup>9</sup>/L) or  $< 35,000/\text{mm}^3$  (35  $\times$  10<sup>9</sup>/L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if due to anemia related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio

- (3 mg/mg or 339 mg/mmol)
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation
- 20. Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) > 2 × the upper limit of normal (ULN) at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK) > 3.0  $\times$  ULN at screening unless related to lupus myositis
- 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic mAb (eg, IgG protein) or molecules made of components of mAbs
- 25. History substance and/or alcohol abuse, or dependence within the past 1 year, at the investigator's judgment
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5

on the Columbia Suicide severity Rating Scale (C-SSRS)

- 31. Current or pending incarceration
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness

#### Statistical Considerations

Below is a summary of the statistical methods. Further details can be found in Section 9.

Baseline and patient characteristics will be summarized via appropriate summary statistics by treatment group and overall, for each phase of the trial.

Binary efficacy endpoints will be compared between treatments via Cochran-Mantel-Haenszel (CMH) analysis. Continuous efficacy endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-by-time interaction, baseline covariate, and covariate-by-time interaction. Summary statistics will be provided by dose/treatment for all safety endpoints. Details will be provided in the statistical analysis plan (SAP).

Two IAs are planned for this study. The initial IA (IA1) will be conducted at the time of the POC decision for dose selection. The second IA (IA2) will be performed for futility. IA2 is planned to be conducted when SRI-4 response is determined for approximately 60 patients (including all patients at the same dose level/matching placebo from the MAD study) after completing 3 months of treatment. The purpose of IA2 is to assess if the trial could stop for an early futility conclusion, or continue. Since there is no plan to stop the trial for an early efficacy conclusion, there is no impact on the type 1 error level.

AEs will be summarized by counts and percentages of patients by treatment group. Laboratory data and vital signs will be summarized by treatment group as summary statistics for value and change from baseline at each individual time point. Summary statistics will include n, arithmetic mean, median, arithmetic SD, minimum, and maximum.

The PK parameter data will be listed and summarized descriptively in tabular format. Binary PD endpoints will be assessed for the full analysis set (FAS) population via CMH analysis. Continuous PD endpoints will be assessed via ANCOVA repeated measures mixed model analysis with multiple factors. PK and PD relationships will be explored graphically and where appropriate model based methods of analysis will used.

# TABLE OF CONTENTS

| TITLE PAGE | 1 |
|----------------------------------------------------|----|
| CLINICAL PROTOCOL APPROVAL FORM | |
| SUMMARY OF CHANGES | 3 |
| CONFIDENTIALITY AND INVESTIGATOR STATEMENT | 17 |
| PROTOCOL SUMMARY | 18 |
| TABLE OF CONTENTS | 31 |
| LIST OF IN-TEXT TABLES | 35 |
| LIST OF IN-TEXT FIGURES | 35 |
| LIST OF ABBREVIATIONS | 36 |
| 1 INTRODUCTION AND RATIONALE | 40 |
| 1.1 Indication | 40 |
| 1.2 Background and Rationale | 40 |
| 1.2.1 Overview of the Disease State | 40 |
| 1.2.2 BOS161721 Development | 40 |
| 1.2.2.1 Interleukin-21 | 41 |
| 1.2.2.2 Preclinical Studies | 42 |
| 1.2.2.3 Clinical Studies | 43 |
| 1.2.3 Study Dose Selection | 44 |
| 1.2.4 Risk-Benefit Assessment | 45 |
| 1.2.5 Potential Risks | 45 |
| 1.2.5.1 Anaphylaxis and Serious Allergic Reactions | 46 |
| 1.2.5.2 Injection Site Reactions | 46 |
| 1.2.5.3 Immune Complex Disease | 47 |
| 1.2.5.4 Infections | |
| 1.2.5.5 Malignancy | 48 |
| 1.2.5.6 Hepatic Function Abnormality | 48 |
| 1.2.5.7 Failure of Vaccination | 49 |
| 1.2.5.8 Potential for Drug-Drug Interactions | 49 |
| 1.2.5.9 Potential Risk to Fetal Development | 49 |
| 2 STUDY OBJECTIVES | 49 |
| 2.1 Phase 1b Multiple Ascending Dose | 49 |
| 2.1.1 Primary Objective | 49 |
| 2.2 Phase 2 Proof of Concept | 50 |
| 2.2.1 Primary Objective | 50 |
| 2.2.2 Secondary Objectives | 50 |
| 3 STUDY ENDPOINTS | 50 |
| 3.1 Phase 1b MAD Study | 50 |
| 3.1.1 Primary Endpoints | 50 |
| 3.1.2 Exploratory Endpoints | 51 |

| 3.1.3 | Other Endpoints | 51 |
|---------|-----------------------------------------------|----|
| 3.1.4 | PRO Endpoints | 52 |
| 3.2 | Phase 2 POC Study | 52 |
| 3.2.1 | Primary Efficacy Endpoint | 52 |
| 3.2.2 | Secondary Efficacy Endpoints | 52 |
| 3.2.3 | Exploratory Endpoints | 53 |
| 3.2.4 | Other Endpoints | 53 |
| 3.2.5 | PRO Endpoints | 53 |
| 4 S | TUDY PLAN | 53 |
| 4.1 | Study Design | 53 |
| 4.1.1 | Multiple Ascending Dose Phase 1b Study | 54 |
| 4.1.1. | Dose Escalation for the MAD Study | 54 |
| 4.1.1.2 | 2 Dose Limiting Toxicity (DLT) | 55 |
| 4.1.1. | 3 DMC Recommendations | 55 |
| 4.1.2 | POC Phase 2 Study | 56 |
| 4.1.2. | 1 BOS161721 Dose | 56 |
| 4.1.2.2 | POC Study Design | 56 |
| 4.2 | Study Schematic | 57 |
| 4.3 | Schedule of Assessments | 58 |
| 5 P | OPULATION | 66 |
| 5.1 | Participant Recruitment | 66 |
| 5.2 | Number of Patients | 66 |
| 5.3 | Patient Screening | 66 |
| 5.4 | Inclusion Criteria | 66 |
| 5.5 | Exclusion Criteria | 68 |
| 5.6 | Concomitant Medications | 70 |
| 5.6.1 | Oral Corticosteroid Dose | 71 |
| 5.6.2 | Other Prohibited and/or Restricted Treatments | 72 |
| 5.7 | Women of Childbearing Potential | 72 |
| 5.7.1 | Determination of Menopause | 72 |
| 5.7.2 | Contraception | 73 |
| 5.8 | Deviation from Inclusion/Exclusion Criteria | 73 |
| 5.8.1 | Patient Withdrawal and Replacement | 74 |
| 6 S | TUDY PROCEDURES | 74 |
| 6.1 | Screening | 74 |
| 6.1.1 | Retesting During Screening Period | 75 |
| 6.2 | Enrollment/Randomization and Day 0 Treatment | 76 |
| 6.3 | Treatment Period/Follow-Up Visits | |
| 6.4 | Safety Follow-Up Visits | |
| 6.5 | Premature Discontinuation | |
| 7 A | ASSESSMENTS | 80 |
| 7.1 | Medical History, Demographic and Other Baseline Information | 80 |
|---------|--------------------------------------------------------------|----|
| 7.2 | Safety Assessments | 81 |
| 7.2.1 | Laboratory Assessments | 81 |
| 7.2.1.1 | Pregnancy testing | 83 |
| 7.2.1.2 | Tuberculosis Screening | 83 |
| 7.2.2 | Adverse Events | 84 |
| 7.2.2.1 | Definitions | 84 |
| 7.2.2.2 | Recording of Adverse Events | 84 |
| 7.2.2.3 | Severity of Adverse Events | 84 |
| 7.2.2.4 | Causality of Adverse Events | 85 |
| 7.2.2.5 | Seriousness of Adverse Events | 85 |
| 7.2.2.6 | Adverse Events of Special Interest | 86 |
| 7.2.2.7 | Reporting of Adverse Events | 89 |
| 7.2.2.8 | Follow Up of Adverse Events | 91 |
| 7.2.3 | Vital Signs | 91 |
| 7.2.4 | 12-Lead Electrocardiograms | 91 |
| 7.2.5 | Physical Examinations | 92 |
| 7.2.6 | C-SSRS | 92 |
| 7.2.7 | Injection Site Reactions | 92 |
| 7.2.8 | Immunogenicity | 92 |
| 7.3 | Efficacy Assessments | 93 |
| 7.3.1 | SLEDAI-2K | 93 |
| 7.3.2 | BILAG 2004 | 93 |
| 7.3.3 | PGA of Disease Activity | 94 |
| 7.3.4 | Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response | 94 |
| 7.3.4.1 | SRI-4 Response | 94 |
| 7.3.4.2 | SRI-5 and SRI-6 Response | 94 |
| 7.3.4.3 | BICLA Response | 94 |
| 7.3.5 | CLASI Response | 95 |
| 7.3.6 | ACR-28 Joint Count | 95 |
| 7.4 | Other Variables | 95 |
| 7.4.1 | SLICC/ACR Damage Index | 95 |
| 7.4.2 | PROs | 95 |
| 7.5 | Pharmacokinetic Assessments | 96 |
| 7.6 | Pharmacodynamic Assessments | 96 |
| 7.7 | Pharmacokinetic/Pharmacodynamic Relationship | 96 |
| 7.8 | Protocol Deviations | 96 |
| 8 ST | TUDY DRUG MANAGEMENT | 97 |
| 8.1 | Description | 97 |
| 8.1.1 | Formulation | |
| 8.1.2 | Storage | 97 |

| 8.2 | Packaging and Shipment | 97 |
|-------------|---------------------------------------------------------|-----|
| 8.3 | Dose and Administration | 97 |
| 8.4 | Accountability | 98 |
| 8.5 | Prohibited Concomitant Therapy | 98 |
| 8.6 | Compliance | |
| 9 S | TATISTICS | |
| 9.1 | Sample Size | 98 |
| 9.2 | Statistical Methods | 99 |
| 9.2.1 | Analysis Populations | 99 |
| 9.2.2 | Demographics and Baseline Characteristics | 99 |
| 9.2.3 | Primary Endpoint(s) | 100 |
| 9.2.4 | Secondary Endpoint(s) | 100 |
| 9.2.5 | Analysis of Safety | 100 |
| 9.2.5. | 1 Safety Analysis | 100 |
| 9.2.5.2 | Data Monitoring Committee | 100 |
| 9.2.6 | Pharmacokinetic and Pharmacodynamic Data | 101 |
| 9.2.6. | 1 Analysis of Pharmacokinetic Data | 101 |
| 9.2.6.2 | 2 Analysis of Pharmacodynamic Data | 101 |
| 9.2.6.3 | Population Pharmacokinetic Analysis or PK/PD Modeling | 101 |
| 9.3 | Interim Analysis and Power | 102 |
| 10 E | THICS AND RESPONSIBILITIES | 102 |
| 10.1 | Good Clinical Practice | 102 |
| 10.2 | DMC | 102 |
| 10.3 | Institutional Review Board/Independent Ethics Committee | 103 |
| 10.4 | Informed Consent. | 103 |
| 10.5 | Records Management | 103 |
| 10.6 | Source Documentation | 104 |
| 10.7 | Study Files and Record Retention. | 104 |
| 11 A | UDITING AND MONITORING | 104 |
| 12 A | MENDMENTS | 105 |
| | TUDY REPORT AND PUBLICATIONS | |
| | TUDY DISCONTINUATION | |
| 15 C | ONFIDENTIALITY | 106 |
| | EFERENCES | |
| 17 A | PPENDICES | |
| <b>APPE</b> | NDIX 1 NAMES OF STUDY PERSONNEL | |
| | NDIX 2 DECLARATION OF HELSINKI | |
| | NDIX 3 COMMONLY USED CORTICOSTEROID EQUIVALENTS | |
| <b>APPE</b> | NDIX 4 MEDICATION WASHOUT PERIODS | |
| <b>APPE</b> | NDIX 5 BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA) | 118 |

# LIST OF IN-TEXT TABLES

| Table 1. | Schodule of Aggaggments Dhogo 1h Multiple Agganding Dage | 50 |
|---|---|---|
| | Schedule of Assessments - Phase 1b - Multiple Ascending Dose | |
| Table 2. | Schedule of Assessments - Phase 2 Proof of Concept (POC) Study | 62 |
| Table 3. | Laboratory Tests | 82 |
| Table 4. | Causality Definitions | 85 |
| Table 5. | Sample Size | 99 |
| | LIST OF IN-TEXT FIGURES | |
| Figure 1. | Individual pSTAT3 C <sub>min</sub> Levels Versus Dose | 44 |
| Figure 2. | Study Diagram for MAD Phase 1b and POC Phase 2 Studies | 57 |

#### LIST OF ABBREVIATIONS

ACR American College of Rheumatology

ADA anti-drug antibody
AE adverse event

AIDS acquired immune deficiency syndrome

ALT alanine aminotransferase ANA antinuclear antibodies ANC absolute neutrophil count

APL antiphospholipid

AST aspartate aminotransferase

AUC area under the concentration-time curve

AZA azathioprine

BICLA BILAG-based Composite Lupus Assessment

BILAG British Isles Lupus Assessment Group

BP blood pressure BUN blood urea nitrogen

BW body weight C complement

C-SSRS Columbia Suicide Severity Rating Scale

CD cluster of differentiation

CK creatine kinase

C<sub>L</sub> systematic clearance

CLASI Cutaneous Lupus Erythematosus Area and Severity Index

C<sub>max</sub> maximum plasma concentration

CMH Cochran-Mantel-Haenszel

CS corticosteroids
CSR clinical study report
DILI drug-induced liver injury
DLT dose-limiting toxicity
DMC data monitoring committee

dsDNA double-stranded deoxyribonucleic acid

ECG electrocardiogram
EOT end of treatment

eCRF electronic case report form

F female

Fc fragment crystallizable

FDA Food and Drug Administration
FSH follicle stimulating hormone

GCP Governor Climical Provides

GCP Good Clinical Practice

eGFR estimated glomerular filtration rate

GLP Good Laboratory Practice

GWAS genome-wide association studies

γc gamma chain HBV hepatitis B virus

hCG human chorionic gonadotropin

HCl hydrochloride HCV hepatitis C virus

HIV human immunodeficiency virus

HR heart rate

HRT hormone replacement therapy

IA interim analysis

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonization

IEC Independent Ethics Committee

Ig immunoglobulin IL interleukin

IL-21R interleukin 21 receptor

IM intramuscular INFγ interferon gamma

INR International Normalized Ratio IRB Institutional Review Board

IUD intrauterine device

IV intravenous

IVRS interactive voice response system

JAK Janus kinase kg kilogram

KLH keyhole limpet hemocyanin LOCF last observation carried forward

M male

mAb monoclonal antibody
MAD multiple ascending dose

MAPK mitogen-activated protein kinase

MS multiple sclerosis MTX methotrexate

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events NIAID/FAAN National Institute of Allergy and Infectious Diseases/Food Allergy and

Anaphylaxis Network

NK natural killer

NOAEL no observed adverse event level

NO nitric oxide

OTC over-the-counter
PD pharmacodynamics
PEF peak expiratory flow

PGA Physician's Global Assessment

PK pharmacokinetics POC proof of concept

PR (interval) from onset of the p-wave to the end of the r-wave

pSS primary Sjögren's syndrome

pSTAT3 phosphorylated signal transducer and activator of transcription 3

PT preferred term

QRS (interval) from the onset of the q-wave to the end of the s-wave
QT (interval) from onset of the QRS complex to the end of the T wave
QTcF QT interval corrected for heart rate using Fridericia's formula

QFT-G QuantiFERON-TB Gold In-Tube

RA rheumatoid arthritis RNP ribonucleoprotein

RR (interval) from the onset of the r-wave to the onset of the next consecutive r-wave

SAD single ascending dose SAE serious adverse event SAP statistical analysis plan

SC subcutaneous

SDMT safety data monitoring board

CCI

SLE systemic lupus erythematosus SLEDAI-2K SLE Disease Activity Index 2000

SLICC Systemic Lupus International Collaborating Clinics

Sm Smith

SOC system organ class
SRI-4 SLE Responder Index 4
SRI-5 SLE Responder Index 5
SRI-6 SLE Responder Index 6
SSA Sjögren syndrome-A (Ro)
SSB Sjögren syndrome-B (La)

STAT3 signal transducer and activator of transcription 3 SUSAR suspected unexpected serious adverse reaction

t<sub>1/2</sub> terminal elimination half-life

TB tuberculosis

TDAR T-cell dependent antibody response

Tfh T-follicular helper

Th T-helper
TK toxicokinetics

Clinical Study Protocol: BOS161721-02

T<sub>max</sub> first time to maximum concentration

Treg regulatory T-cell TT tetanus toxoid

ULN upper limit of normal

US United States

Vd volume of distribution

WBC white blood cell

WHO World Health Organization
WOCBP women of childbearing potential

YTE triple mutation

#### 1 INTRODUCTION AND RATIONALE

#### 1.1 Indication

BOS161721 is a humanized monoclonal antibody (mAb), which binds to and inhibits interleukin-21 (IL-21) bioactivity, and is being developed for the treatment of moderately to severely active systemic lupus erythematosus (SLE) in adults.

# **1.2** Background and Rationale

#### 1.2.1 Overview of the Disease State

SLE is a chronic inflammatory autoimmune disease that has variable manifestations in multiple organ systems and follows a relapsing and remitting course. The disease process includes abnormal immune responses mediated by tissue-binding autoantibodies and immune complex deposition, giving rise to tissue damage often resulting in end organ disease and even mortality. Survival of SLE has improved due to earlier detection, improved overall medical care, and standardized SLE treatment with corticosteroids, immunosuppressants, and cytotoxic agents. However, some of the morbidity in patients with SLE is related to its treatment. Comparison of early and late outcomes in patients with SLE demonstrate that death in early disease is most commonly due to infections and active SLE causing multi-system organ damage, while thromboses were the most common cause of death during later disease.<sup>2</sup>

The reported prevalence of SLE in the United States (US) is 20 to 70 cases per 100,000 people.<sup>3</sup> More than 90% of cases of SLE occur in women, frequently starting at childbearing age. Women of color are disproportionately affected by SLE. This suggests multiple genetic and environmental factors are at play. Accordingly, a multifactorial view of the immunopathogenesis of SLE suggests more than 1 area of interest, including breach in central tolerance in the adaptive arm of the immune system, peripheral amplification of the autoimmune response by the innate immune system, and local processes in the target organ that facilitate end-organ disease.<sup>4</sup>

#### **1.2.2 BOS161721 Development**

Boston Pharmaceuticals is developing BOS161721 for the treatment of SLE. BOS161721 is a humanized immunoglobulin G1 (IgG1) mAb directed against human IL-21.

Murine mAb 19E3, the progenitor of BOS161721, was generated using mouse hybridoma technology. 19E3 has subpicomolar (pM) affinity to human IL-21 and was selected for its potent neutralization of IL-21 bioactivity. BOS161721 was generated by the humanization of mAb 19E3 where its complementarity-determining regions were grafted onto a human IgG1 kappa backbone. The fragment crystallizable (Fc) portion of BOS161721 contains a YTE (M252Y/S254T/T256E triple mutation) in the constant domain of the IgG1 heavy chain that was introduced into the parental molecule, 19E3, intended to prolong the in vivo terminal elimination half-life (t<sub>1/2</sub>) of the mAb.<sup>5</sup> Thus, BOS161721 retains sub-pM binding to IL-21 and prevents IL-21 from binding to the IL-21 receptor (IL-21R), inhibiting IL-21 bioactivity.

BOS161721 binds to human IL-21 and Cynomolgus monkey IL-21, which are highly homologous, and neutralizes the bioactivity of both. BOS161721 is specific for IL-21 as it does not bind to or inhibit the other gamma-chain (γc) family of cytokines, and acts to specifically neutralize the IL-21 pathway. In *in vitro* studies, BOS161721 inhibited downstream IL-21-induced signaling, IL-21-induced plasma cell differentiation, and IL-21-induced natural killer (NK) cell activation. In *in vivo* studies, BOS161721 significantly inhibited the T-cell dependent antibody response (TDAR) to immunization with a protein antigen as well as B-cell expansion following a second protein antigen immunization in Cynomolgus monkeys.

#### **1.2.2.1** Interleukin-21

IL-21 is an inflammatory cytokine, which belongs to a family of cytokines that also includes IL-2, IL-4, IL-7, IL-9, and IL-15, all of which bind to private receptors in complex with the common cytokine receptor yc. Most cytokines in this family are critically important for both the maintenance and function of T-cell and B-cell responses. IL-21 signals through a receptor complex consisting of its own private receptor, the IL-21R and vc. 6,7 Engagement of the IL-21R/γc complex leads to the activation of several signaling pathways, including the Janus kinase/signal transducer and activator of transcription, mitogen-activated protein kinase (MAPK) and phosphoinositide 3-kinase pathways.<sup>8</sup> IL-21 is produced mainly by T-cells and NK T-cells, but neutrophils have also been reported to produce IL-21. 9,10 The IL-21R is expressed on a broad array of cell types, including B-cells, T-cells, NK-cells, macrophages and dendritic cells, as well as other hematopoietic and nonhematopoietic cells such as fibroblasts, keratinocytes, and intestinal epithelial cells. 9,11 Activation of signal transducer and activator of transcription 3 (STAT3) via phosphorylation is critical in regulating human B-cell responses to IL-21<sup>12</sup>; phosphorylated STAT3 (pSTAT3) forms a homodimer, which translocates to the nucleus where it initiates transcription of the IL-21 gene, forming an autocrine loop for IL-21 production via STAT3 phosphorylation. <sup>13</sup> In addition, IL-21 has been shown to upregulate expression of its own receptor <sup>14</sup> and induces an autocrine feedback loop. <sup>15</sup>

IL-21 modulates various aspects of immune function. It promotes cluster of differentiation 4 (CD4+) T-cell differentiation and promotes the generation of T-helper (Th)17<sup>16</sup> and T-follicular helper (Tfh) cells. <sup>15,17</sup> In mice, IL-21 has been shown to regulate the balance between Th17 and regulatory T-cell (Treg), in that it increases Th17, while inhibiting Treg differentiation. <sup>18</sup> Less is understood with regards to human Tregs, although IL-21 has been reported to counteract Treg suppression of human effector T-cells and blockade of IL-21 promotes Treg generation in a murine model of graft versus host disease induced by human T-cells. <sup>20</sup> IL-21 upregulates CD8+ T-cell and NK-cell expansion and cytolytic activity by increasing granzyme B and perforin. <sup>21,22</sup> IL-21 also has been reported to increase granzyme B in plasmacytoid dendritic cells and B-cells resulting in inhibition of T-cell responses. <sup>23,24</sup> IL-21 also has a variety of effects on nonhematopoietic cells, such as stromal cells and induces inflammation through matrix metalloproteinase release by gut intestinal fibroblasts. <sup>25</sup>

One principal non-redundant role of IL-21 is the promotion of B-cell activation, differentiation, or death during humoral immune responses. <sup>14</sup> Furthermore, increased IL-21 production is characteristic of several autoimmune diseases and is likely to contribute to autoantibody production as well as pathologic features of autoimmune disease. <sup>26</sup> The critical role of IL-21 in promoting humoral and other immune responses makes it an important focus of potential

therapeutic interventions in conditions characterized by overproduction of pathogenic autoantibodies. IL-21 production by Tfh cells in humans is believed to play a major role in driving the autoantibody production through its role in plasma cell differentiation. Importantly, Tfh cell populations are expanded in patients with autoimmune diseases such as lupus, bullous pemphigoid, rheumatoid arthritis (RA) and primary Sjögren's syndrome (pSS) and have been reported to correlate with IL-21 levels, autoantibodies, and disease severity. <sup>26,27,28,29</sup> Furthermore, loss of number and functionality of Tregs has been associated with autoimmune diseases such as SLE and giant cell arteritis, which IL-21 is expected to modulate. <sup>30,31</sup> Thus, neutralization of IL-21 in settings of autoimmunity is expected to impact several cell populations believed to be involved in the pathogenesis of autoimmune disorders including SLE.

BOS161721 selectively binds IL-21 with high affinity to neutralize IL-21, and due to its pleiotropic nature, neutralization of IL-21 is expected to impact several cell populations believed to be involved in the pathogenesis of SLE. Importantly, patients with SLE have elevated IL-21 plasma levels that correlate with the severity of the disease. Recently, genome-wide association studies (GWAS) have provided convincing evidence that the chromosomal 4q 27 region harbors the IL-21 genes and is associated with chronic inflammatory disorders, including SLE.<sup>29</sup>

#### 1.2.2.2 Preclinical Studies

The pharmacokinetics (PK) of BOS161721 were characterized following single-dose intravenous (IV) administration of BOS161721 (0.01 to 30 mg/kg) in male Cynomolgus monkeys or repeat, every 2 weeks IV administration (15 to 100 mg/kg) and subcutaneous (SC) administration (50 mg/kg) in male and female Cynomolgus monkeys. Systemic exposure was approximately dose-proportional within the tested dose range. SC bioavailability was determined to be 64.3%.

Two single-dose (IV) non-good laboratory practice (GLP) studies conducted in Cynomolgus monkeys evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), and immunogenicity of BOS161721. Following a single IV administration (slow bolus), there were no BOS161721-related adverse changes, resulting in a no-observed-adverse-effect-level (NOAEL) value of 30 mg/kg, the highest dose tested among 2 studies.

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) administration for 3 months (a total of 7 doses).



#### 1.2.2.3 Clinical Studies

BOS161721-01 was a double-blind, Phase 1, single ascending dose (SAD) study to assess the safety, PK, and PD of BOS161721 in healthy subjects. The primary objective of the study was to characterize the safety and tolerability of IV and SC SADs of BOS161721 in an otherwise healthy subject population without concomitant illnesses, immune abnormalities, or concomitant medications. Secondary objectives included characterization of the PK and immunogenicity of BOS161721, and exploratory objectives included the evaluation of the effect of BOS161721 on TDAR to keyhole limpet hemocyanin (KLH) (primary and secondary immunizations) in healthy subjects, the effects of BOS161721 on plasma levels of IL-21 (free and bound), and the evaluation of the effect of BOS161721 on IL-21 gene expression (via gene signature) in blood. This study consisted of 8 cohorts. Subjects were randomized in a 3:1 ratio (BOS161721: placebo) and received either a single dose of BOS161721 (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) or placebo, with safety follow-up. For the first cohort, after the first 2 subjects were dosed (1 active and 1 placebo), there was a minimum gap of 48 hours before the remaining subjects from that cohort were dosed, to allow for an initial review of any emerging safety and tolerability data. For all cohorts, escalation to the next dose was not sooner than 8 days after all the subjects in the prior cohort had been dosed and were based on a review of at least 7 days of safety and tolerability data by the Safety Data Monitoring Team (SDMT).

Blood samples were collected at every in-house study visit for BOS161721 concentration determinations. Blood samples were also collected for determination of IL-21 plasma levels (free and total). Safety was assessed based on the occurrence of treatment-emergent AEs, hepatic function abnormality, and acute and delayed hypersensitivity reactions. Other safety variables included electrocardiograms (ECGs), vital signs (blood pressure, heart rate, and temperature), safety laboratory assessments, blood sampling for ADAs, total IgG and IgM levels, CD4+ count, and full and targeted physical examinations. Overall, there were no clinically significant findings from this study, following an interim cut and review of the data at Day 90 postdose. Adverse events reported as related to the study drug, particularly infections, were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. There was 1 serious adverse event (SAE; death due to pulmonary embolism) that occurred 127 days after a single administration of 240 mg SC dose of BOS161721. The causality of this single SAE was not attributed to study drug and further information can be found in the Investigator's Brochure. PK data from the SAD study demonstrates BOS161721 has an extended  $t_{1/2}$  (provisional single dose data indicates this to be approximately 42-46 days) which supports evaluation of monthly dosing.

### 1.2.3 Study Dose Selection

Doses have been selected for the multiple ascending dose (MAD) Phase 1 study based on a 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01); the SDMT reviewed the blinded safety data from subjects for each dose cohort (8 cohorts, evaluating 1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg), along with the accumulated safety and available PK/PD data from all subjects in the previous dose cohorts, to make a decision on whether to proceed to the next higher dose level, repeat a dose level, or stop dose escalation. Overall, there were no clinically significant safety or tolerability findings from this study.

Based on the Day-90 interim cut of the PK and biomarker data in the BOS161721-01 study, the recommended doses for evaluation in the MAD phase of this study are 20, 60, and 120 mg SC monthly. This dose recommendation is supported by evidence of linear PK with BOS161721 resulting in a median  $T_{max}$  of 6 days and an apparent terminal half-life of 44 days. Furthermore, pSTAT3 suppression, a marker of IL-21 target engagement, follows a similar time course of the mAb levels, with maximal and sustained suppression apparent with doses greater than 30 mg SC (Figure 1).



Figure 1. Individual pSTAT3 C<sub>min</sub> Levels Versus Dose

IV = intravenous, pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SC = subcutaneous

All doses selected for the MAD study are projected not to exceed the mean exposure of that achieved following the highest single dose of 240 mg SC administered in the Phase 1 SAD study. Cohort 1 will include randomized treatment to the 20 mg dose. Based on the staggered study design, the data monitoring committee (DMC) will perform a scheduled review of safety data and sequentially consider dose escalation for Cohorts 2 and 3. In addition, the DMC and Boston Pharmaceuticals will conduct a data review for the first interim analysis (IA1). At that time, a decision will be made to suggest which dose should be carried forward into the proof of concept (POC) Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD study (see Section 4.1.1.1).

#### 1.2.4 Risk-Benefit Assessment

The available preclinical data on BOS161721, the findings in clinical study BOS161721-01, and existing clinical information on IL-21 inhibitors suggest that the present clinical study has an acceptable risk-benefit ratio. In this study, the risk-benefit assessment of BOS161721 in adult patients with moderately to severely active SLE will be ongoing, with step-wise evaluations during the staggered MAD study. The DMC used in this study is charged with assessing such actions in light of an acceptable benefit-risk profile for BOS161721 as an anti-IL-21 mAb. Formal DMC monitoring meetings will occur as described in the DMC Charter. Two weeks after Cohort 1 has received a second dose of study drug, the DMC will evaluate the safety and tolerability data from Cohort 1 to determine the recommended dose for Cohort 2. Two weeks after 8 patients in Cohort 2 receive a second dose, the DMC will determine if dose escalation to Cohort 3 can proceed. Two weeks after the last patient in Cohort 3 receives the second dose, the DMC and Boston Pharmaceuticals will conduct a data review for the IA1. At that time, a decision will be made to suggest which dose should be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of doselimiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 during the MAD study. Thereafter, DMC monitoring will be conducted periodically throughout the study as described in the DMC charter. With the agreement of the DMC and sponsor, this schedule may be modified depending on the rate of patient accrual. Additional details can be found in the DMC Charter.

The benefit of participation for all patients in this study is close monitoring of their medical condition and safety of their treatment. Those randomized to the active treatment arm may potentially experience improvement in their SLE disease. Those randomized to the placebo (in combination with standard of care) arm are not expected to obtain any additional benefit, beyond those of their background treatment, though close monitoring of their medical condition and safety may itself be associated with improving their SLE.

#### 1.2.5 Potential Risks

Potential risks based on the mechanism of action of BOS161721 include infections, risks associated with the administration of any foreign protein or biologic agent, including injection site reaction, anaphylaxis, serious allergic reaction, and development of ADAs. ADAs could result in immune complex disease (with manifestations such as arthralgias, serum-sickness, and vasculitis), autoimmunity, or altered BOS161721 levels or activity. Further details can be found

in the current Investigator's Brochure (IB) for BOS161721, which contains comprehensive toxicology, preclinical and clinical information on BOS161721.

Two investigational drug products are considered to be in the same pharmacological class as BOS161721 based on interruption of signaling through the IL-21 signaling pathway. No potential risk generalizable across the class has been observed with these investigational products. Based on the clinical Phase 1 SAD study (BOS161721-01), AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs.

The majority of IgG elimination occurs via intracellular catabolism, following fluid-phase or receptor-mediated endocytosis. This type of endocytosis and elimination is a form of target-mediated disposition where the interaction of the drug and its pharmacological target (eg, a target receptor) serves as a significant contributor to the kinetics of antibody distribution and elimination. Renal elimination, which is a primary pathway of clearance of small-molecule drugs, is relatively unimportant for IgG, as its large size prevents efficient filtration through the glomerulus. Secretion into the bile is an important pathway of elimination of IgA antibodies, but this route is not a significant contributor to the elimination of IgG antibodies. Thus, risk to renal and hepatic systems due to metabolism of BOS161721 is low.<sup>33</sup>

### 1.2.5.1 Anaphylaxis and Serious Allergic Reactions

As with the administration of any foreign protein and/or other biological agents, acute hypersensitivity reactions, including acute anaphylactic/hypersensitivity, severe allergic, and anaphylactoid reactions may follow infusion of mAbs and can be caused by various mechanisms. These acute hypersensitivity reactions may be severe and result in death.

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria,<sup>34</sup> and are discussed in Section 7.2.2.6.1.

Based on the limited Phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed.

Patients with a known history of allergy or severe hypersensitivity reaction to any component of BOS161721 formulation or patients with a history of anaphylaxis to any other biological therapy such as mAbs will be excluded from studies with BOS161721. In addition, appropriate drugs and medical equipment to treat acute hypotensive, bronchoconstrictive, or anaphylactic reactions will be immediately available at the unit and study personnel will be trained to recognize and treat these reactions.

#### 1.2.5.2 Injection Site Reactions

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) for 3 months (a total of 7 doses); no SC animals had injection reactions.

Based on the Phase 1 SAD study (BOS161721-01), incidence of injection site reactions in subjects who received BOS161721 was similar to placebo.

Patients will be monitored for local injection site reactions in this study. See Section 7.2.7.

#### 1.2.5.3 Immune Complex Disease

The potential risk of immune complex disease for BOS161721 is theoretical, based on the known risks associated with mAbs. The administration of a mAb can result in the formation of ADAs. Administration of the mAb in the presence of ADA may result in the formation of circulating antibody-antigen complexes potentially resulting in altered BOS161721 levels or activity or deposition of the complexes in microvasculature. Complement is frequently involved in the latter setting, and the breakdown products of complement attract polymorphonuclear leukocytes to the site of deposition where they can provoke local tissue damage through specific or nonspecific release of enzymes. Two of the more common end-organ targets are the blood vessels (vasculitis) and kidney (nephritis). These clinical manifestations represent immune complex disease or Type III hypersensitivity. Although BOS161721 is a humanized mAb, ADAs may develop; however, the likelihood of occurrence of immune complex disease with BOS161721 is low. The findings of immune complex disease are typically reversible when mAb administration stops and the antibody-antigen complexes are cleared from the body.

Based on the limited Phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed.

#### 1.2.5.4 Infections

BOS161721 is expected to diminish the activity of T-cell, B-cell and NK-cell lines. Like other medications modulating immune response, BOS161721 may increase the potential risk for infection, including serious infections. IL-21 produced by CD4+ Th cells is required to sustain the anti-viral function of CD8+ T-cells against chronic viral infections. Nonclinical evidence suggests that the risk of chronic viral infection recurrence or increased severity may occur with IL-21 inhibition.<sup>35</sup>

These conditions will be fully characterized with clinical descriptions and routine laboratory and/or specialty testing and treated where indicated with appropriate local standard of care.

Patients with a history of opportunistic infection, including recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years, or any other underlying pathology predisposing to serious infection, are excluded from studies with BOS161721 (for further details please refer to the current IB for BOS161721).

Patients will be assessed for hepatitis B, and C, and HIV-1/2 combination, at screening.

### <u>Cryptosporidium Infection</u>

Cryptosporidium infection was noted in patients with an IL-21 receptor loss-of-function gene mutation and similar findings of cryptosporidium infection have been observed in immunosuppressed liver transplant and human immunodeficiency virus patients. Since

BOS161721 is expected to diminish the immunosurveillance activity of T-cell, B-cell, and NK-cell lines, a similar risk is biologically plausible with prolonged exposure to BOS161721.

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells,<sup>37</sup> patients with a CD4+ count < 500 cell/mm<sup>3</sup> were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from the proposed MAD/POC studies. Patients exposed to investigational product who develop diarrhea during the course of the study should immediately undergo an assessment for opportunistic infection including stool for ova and parasites and stool examination for cryptosporidium. Positive cryptosporidium in stool sample at screening is an exclusion. Treatment by the investigator where indicated should be guided by findings and be consistent with local standard of care.

Based on the limited Phase 1 SAD study (BOS161721-01), infections in subjects who received BOS161721 was not observed.

# 1.2.5.5 Malignancy

The stimulatory effect of IL-21 on NK cells and CD8+ T-cells suggests the cytokine may have anti-tumor activity. Nonclinical studies have demonstrated significant anti-tumor effects of IL-21 in a number of tumor models. IL-21 therapy of human metastatic melanoma and renal cell carcinoma has demonstrated POC with significant increases in levels of perforin, granzyme B, and interferon gamma (IFNγ) expression in CD8+ T-cells and NK T-cells. Clinical response has been limited in these generally unmanageable diseases.

The impact of treatment with anti-IL-21 therapy on the development or growth of malignancies is not known; however, as with other immunomodulatory biologic agents, treatment with BOS161721 may result in an increase in the risk of malignancies. NK cell suppression by IL-21 neutralization may represent a biological mechanism for a potential risk for malignancy. Patients with a history or current diagnosis of cancer within the past 5 years, with the exception of non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy, are excluded from the study.

Based on the limited Phase 1 SAD study (BOS161721-01), malignancy in subjects who received BOS161721 was not observed.

#### **1.2.5.6** Hepatic Function Abnormality

There is no substantial evidence suggesting BOS161721 is associated with liver function abnormality. However, as a precaution, patients with a history of abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST > 2 × upper limit of normal [ULN]; total bilirubin > 1.5 × [ULN] and judged by the investigator to be clinically significant) were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from the MAD study. Patients with a positive hepatitis B or C test or a history of alcohol dependence will also be excluded.

Based on the limited Phase 1 SAD study (BOS161721-01), hepatic function abnormality in subjects who received BOS161721 was not observed.

#### 1.2.5.7 Failure of Vaccination

IL-21 is a key cytokine in development of B-cells into immunoglobulin-secreting plasma cells. Abnormal signaling through the IL-21R/Janus Kinase (JAK)3/signal transducer and activator of transcription (STAT3) pathway leads to defective humoral immune responses to both T-dependent and T-independent antigens and impairs the establishment of long-lasting B-cell memory. Abnormal signaling through the pathway has been related to decreased specific antibody responses following vaccination, and to increased susceptibility to encapsulated bacterial infections.<sup>38</sup>

The effect of BOS161721 was evaluated in in vivo single dose studies in Cynomolgus monkey in which the animals received vaccination to T-cell dependent KLH antigen to stimulate a TDAR. These in vivo studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen; however, it is worth noting that BOS161721 administration did not produce any remarkable changes in anti-KLH antibody data for IgM, IgG1, IgG3, and IgG4 or anti-tetanus toxoid (TT) antibody data for IgM, IgG, IgG1, or IgE during the dosing phase in the same study.

### 1.2.5.8 Potential for Drug-Drug Interactions

Drug-drug interactions were not evaluated in the Phase 1 SAD study (BOS161721-01), which included only healthy adult subjects. Use of prescription medications (with the exceptions of oral contraceptives), and over-the-counter (OTC) treatments including herbal supplements such as St John's Wort (except multivitamins), in the 2 weeks prior to screening was prohibited in the SAD study.

See Section 5.5 for other specific exclusion criteria which support lowered risk of interactions, and Section 5.6.1 for corticosteroid (CS) dosing. In addition, Section 1.2.5.6 describes considerations for hepatic function for this study.

#### 1.2.5.9 Potential Risk to Fetal Development

No data on preclinical reproductive toxicity are available at the time of this study.

#### 2 STUDY OBJECTIVES

This trial has separate primary and secondary objectives for the MAD Phase 1b and POC Phase 2 studies.

# 2.1 Phase 1b Multiple Ascending Dose

# 2.1.1 Primary Objective

To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20 mg, 60 mg, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose.

# 2.2 Phase 2 Proof of Concept

# 2.2.1 Primary Objective

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on the SLE Responder Index 4 (SRI-4), with sustained reduction of oral CS, in adult patients with moderately to severely active SLE on limited background standard of care treatment.

### 2.2.2 Secondary Objectives

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment, including:

- Changes in SLE-specific autoantibody titers
- Changes in complement 3 and 4 (C3 and C4) levels
- Responses on SRI-4, SRI-5, and SRI-6, with sustained reduction of oral CS
- Response on the British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (BICLA)
- Response on the Cutaneous Lupus Erythematosus Area and Severity Index (CLASI)
- Changes in the SLE Disease Activity Index 2000 (SLEDAI-2K)
- Changes in American College of Rheumatology (ACR)-28 joint count

### 3 STUDY ENDPOINTS

This trial has separate primary and secondary endpoints for the MAD Phase 1b and POC Phase 2 studies.

# 3.1 Phase 1b MAD Study

### 3.1.1 Primary Endpoints

Evaluation of safety, tolerability, and immunogenicity at each dose level, to determine the optimal dose, will include the recording of the following parameters:

- Incidence and severity of AEs, AEs of special interest, and SAEs
- 12-lead ECGs
- Vital signs (blood pressure [BP], heart rate, and temperature)

- Clinical laboratory assessments
- Physical examinations
- Evaluation for ADAs

# 3.1.2 Exploratory Endpoints



# 3.1.4 PRO Endpoints

• CCI

• CCI

### 3.2 Phase 2 POC Study

### 3.2.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the proportion of patients who achieve treatment response as measured by the SRI-4 at Day 210, along with a sustained reduction of oral CS ( $\leq$  10 mg/day and  $\leq$  Day 0 dose) between Day 120 and Day 210

### 3.2.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints are:

- The proportion of patients who achieve treatment response for the SRI-5 and SRI-6 at Day 210, along with a sustained reduction of oral CS (≤ 10 mg/day and ≤ Day 0 dose) between Day 120 and Day 210
- Changes from baseline in dsDNA, ANA, SSA, SSB, RNP, Sm, APL autoantibodies, at Day 120 and Day 210
- Changes from baseline in C3 and C4 levels at Day 120 and Day 210
- Changes from baseline in the SLEDAI-2K at Day 210
- Time to BILAG A or B flare
- Changes from baseline in the CLASI at Day 210
- The proportion of patients with a BICLA response at Day 210
- The proportion of patients with CLASI response at Day 210
- Changes from baseline (percentage) in swollen joints and tender joints ACR-28 joint count
- Incidence and severity of AEs, AEs of special interest, and SAEs
- 12-lead ECGs
- Vital signs (BP, heart rate, and temperature)
- Clinical laboratory assessments

- Physical examinations and targeted physical examinations
- Evaluation for ADAs

# 3.2.3 Exploratory Endpoints



# 4 STUDY PLAN

# 4.1 Study Design

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of SC doses of BOS161721 in adult patients with

moderately to severely active SLE. After successfully completing a screening phase, patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly.

The trial will consist of 2 studies: MAD Phase 1b, and POC Phase 2. Both studies will be double-blinded, and patients will have the same number of visits. Patients may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180, followed by a 90-day safety follow-up visit.

SLE disease activity assessment data will be centrally reviewed by medical monitor and sponsor to ensure the scores are clinically meaningful and compliant with specific definition. The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease being studied. Further details on the content and methods of data reports by the medical monitor and sponsor will be outlined in the Medical Data Review Plan along with the processes and procedures that will be followed.

# 4.1.1 Multiple Ascending Dose Phase 1b Study

The MAD study will consist of 3 cohorts:

- Cohort 1 (20 mg SC) will include 6 patients
  - o 5 patients will receive BOS161721 (active group) and 1 patient will receive placebo (placebo group)
- Cohorts 2 (60 mg SC) and 3 (120 mg SC) will include 12 patients each
  - o 9 patients in the active group and 3 in the placebo group

Doses selected for each of the 3 cohorts is based on a 90-day safety, tolerability, PK and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. All doses selected for the MAD study are projected not to exceed the mean exposure of that achieved in the SAD study.

#### 4.1.1.1 Dose Escalation for the MAD Study

The MAD study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after DMC evaluation of the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing after DMC evaluation of the safety and tolerability data from Cohorts 1 and 2. Each cohort will continue at their assigned dose level through their respective 6-month treatment periods (See Study Schematic, Section 4.1). If > 3 patients discontinue the study in a cohort, he/she may be replaced.

Criteria for dose escalation are further described in the DMC Charter. See Section 4.1.1.2 for additional details about DLTs.

#### **4.1.1.2 Dose Limiting Toxicity (DLT)**

Severity of adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs occurring after study drug administration, which are attributable to the study drug, will be considered DLTs:

#### **Hematologic:**

- Grade 4 neutropenia
- Grade 3 neutropenic infection
- Grade 3 thrombocytopenia with bleeding
- Grade 4 thrombocytopenia

### **Non-Hematologic:**

- Grade 3 or above toxicities, persisting after optimal treatment with standard medical therapy (eg, anti-emetics, anti-diarrheals)
- Drug-induced liver injury ([DILI], Hy's Law), as defined in Section 7.2.2.6.3

Investigators should always manage their patients according to their medical judgment which may include interruption of study drug based on the particular clinical circumstances.

#### 4.1.1.3 DMC Recommendations

During scheduled meetings, the DMC will review relevant study data for safety or benefit-risk concern. During the MAD study, the DMC may provide the following recommendations to the sponsor:

- Expanding a cohort at a specific dosing level, or repeating a lower dose in a subsequent cohort
- Continuing a dose level for a given cohort
- Escalating a dose level for a subsequent cohort
- Termination of current or previous cohort(s)

Further dosing in a given cohort will be halted if 2 or more DLTs are identified intra- and inter-patients dosed. For the POC study, the DMC and Boston Pharmaceuticals will conduct a data review for the IA1 to suggest which dose should be carried forward into the POC Phase 2

study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available at the time the last patient in Cohort 3 completes the Day 44 visit (2 weeks after dose 2). Details are provided in the DMC Charter.

### 4.1.2 POC Phase 2 Study

#### 4.1.2.1 BOS161721 Dose

The optimal dose evaluation is chosen based on MAD Phase 1b safety, tolerability, immunogenicity, and PK and PD data. The dose will be communicated by a letter to site investigators participating in the POC Phase 2 study, and to the IRB/IEC.

# 4.1.2.2 POC Study Design

For the POC study, approximately 156 patients will be randomized to active or placebo groups in a 2:1 ratio.

As in the MAD study, each patient in the POC study may receive a total of 7 SC monthly doses of study drug on Days 0, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Section 4.3). Dose selection will be based on the sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD study of 30 patients treated with BOS161721/placebo.

Data from approximately 60 patients (including the 12 from the MAD study, or 6 fewer if the low dose is chosen who are in the cohort of the chosen dose for the POC study) who complete 3 months of treatment will be used in the IA2 at Day 90 to assess if the trial could stop for an early futility conclusion (see Section 9.3 for details regarding the IA). If futility is not claimed in the IA2, the POC study will continue to approximately 156 patients.

Following the 6-month treatment period, primary and secondary efficacy endpoints will be assessed for each patient after providing their Day 180 disease activity assessments.

DMC monitoring will be conducted periodically throughout the study as described in the DMC charter.

BOS161721 Boston Pharmaceuticals, Inc. Clinical Study Protocol: BOS161721-02

# 4.2 Study Schematic

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2 Studies



A = active drug (BOS161721); P = placebo


### Clinical Study Protocol: BOS161721-02

**Schedule of Assessments** 

4.3

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | | | Safet | y Follov | v-Up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| GENERAL ASSESSM | 1ENTS | | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| SLICC Criteria for<br>SLE | X | | | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>c</sup> | | X | | | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | | X | | X | X | X | X | X | | | | | |
| SAFETY ASSESSME | NTS | | • | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | | | |
| Chest x-ray <sup>d</sup> | X | | | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>e</sup> | X | X | | | X | | | X | | | | | | | | X |
| Injection site reaction assessment <sup>f</sup> | | X | X | | X | | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | | X | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>g</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESSM | MENTS | | | | | | | | | | | | | | | |
| BILAG-2004 Index | X | X | | | X | | X | X | X | X | X | | | X | X | X |


Clinical Study Protocol: BOS161721-02

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | | | | | | | | | | | y Follov | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | - | | 11 | 12 | 13 |
| SLEDAI-2K | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| PGA of disease | | | | | | | | | | | | | | | | |
| activity | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLICC/ACR Damage | | | | | | | | | | | | | | | | |
| Index | | X | | | | | | | | | X | | | | | |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| LABORATORY ASS | ESSMENT | ΓS | | | | | | | | | | | | | | |
| CD4+ count | X | X | | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments | | | | | | | | | | | | | | | | |
| (hematology and | | | | | | | | | | | | | | | | |
| clinical chemistry) <sup>h</sup> | X | X | | | X | X | X | X | X | X | X | | | X | X | X |
| Coomb's test directi | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | | X | X | X | | X | | | X | | | | | |
| Plasma CCI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Plasma CCI & | X | X | | X | X | | X | X | | | X | | | | | |
| Whole blood for | Λ | Λ | | Λ | Λ | | Λ | Λ | | | Λ | | | | | |
| leukocyte | | | | | | | | | | | | | | | | |
| immunophenotype | X | X | | X | X | | X | X | | | X | | | | | |
| ADA <sup>j</sup> | | X | | X | X | | X | X | | | X | | | | | X |
| nAb <sup>k</sup> | | | | | | | | X | | | X | | | | | |
| pSTAT3 | | X | | | X | X | X | X | | | X | | | | | X |
| CCI | | X | | | | | | | | | X | | | | | |
| Whole blood RNA | | 21 | | | | | | | | | 11 | | | | | |
| collection | | X | | X | X | | | X | | | | | | | | X |


Clinical Study Protocol: BOS161721-02

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | Treatment Period Follow-Up 7 | | | | | | | | | | | | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | -28<br>to -1 | 0 | 7<br>(± 1) | 15<br>(± 3) | 30<br>(± 3) | 44<br>(± 3) | 60<br>(± 3) | 90<br>(± 3) | 120<br>(± 3) | 150<br>(± 3) | 180<br>(± 3) | 187<br>(± 3) | 195<br>(± 3) | 210<br>(± 3) | 240<br>(± 3) | 270<br>(± 3) |
| Visit Number | 1 | 2 | - | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| CCI | X | X | | | X | | X | X | X | X | X | | | X <sup>l</sup> | X <sup>1</sup> | X <sup>l</sup> |
| CRP | X | | | | | | | X | | | | | | | | X |
| Serum pregnancy test (women) | X | | | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>m</sup> | | X | | | X | | X | X | X | X | X | | | | | |
| TB test<br>(QuantiFERON-TB<br>Gold In-Tube) <sup>d</sup> | X | | | | | | | | | | | | | | | |
| Serology (hepatitis B and C, HIV-1/2 combination) | X | | | | | | | | | | | | | | | |
| Stool sample <sup>n</sup> | X | | | | | | | | | | | | | | | |
| Spot urine for protein/creatinine ratio | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| PK Labs | | | | | | | | | | | | | | | | |
| Predose <sup>o</sup> | | X | | | X | | X | X | X | X | X | | | | | |
| Postdose | | X <sup>p</sup> | X | X | X <sup>p</sup> | | | | | | X <sup>p</sup> | X | X | X | X | X |


Clinical Study Protocol: BOS161721-02

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screena | Enroll | | | | Tre | atment | Period ! | Follow- | Up | | | | Safet | y Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 7 | 15 30 44 60 90 120 150 180 187 195 | | | | | | | | | | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | (±3) |
| Visit Number | 1 | 2 | - | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | - | - | 11 | 12 | 13 |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; GC ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index;

CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram;

; FSH = follicle stimulating hormone; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G;

IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; nAb = neutralizing antibody; PGA = Physician's Global Assessment;

PK = pharmacokinetic; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; RNA = ribonucleic acid; RNP = ribonucleoprotein;

SAE = serious adverse event; SC = subcutaneous; CC | SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus

International Collaborating Clinics; CC

; TB = tuberculosis; TDAR = T-cell dependent antigen response.

- <sup>a</sup> Screening assessments will be performed over more than 1 visit.
- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 5.6.1 for further details.
- <sup>c</sup> Randomization should occur after patient eligibility has been confirmed by central eligibility review.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- <sup>c</sup> ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed predose and at 2 hours postdose.
- Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 7, 187, and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.
- h Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.
- When clinically indicated.
- Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.
- <sup>k</sup> nAb is assessed if patient is positive for ADA.
- Only dsDNA collected during safety follow-up visits.
- <sup>m</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- <sup>n</sup> Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- <sup>o</sup> Predose samples occur on study drug administration visit days.
- Postdose samples will be collected at 4, 8, and 24 hours after study drug administration on Days 0, 30, and 180.


Clinical Study Protocol: BOS161721-02

Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screen | Enroll | | | | Safe | ty Follo | w-Up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | | 10 | 11 | 12 |
| GENERAL ASSESSMENTS | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| SLICC Criteria for SLE | X | | | | | | | | | | | | | |
| Concomitant medication <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization <sup>c</sup> | | X | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | X | X | X | X | X | X | | | | | |
| SAFETY ASSESSMENTS | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | |
| Chest x-ray <sup>d</sup> | X | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | X | | | X | | | | | |
| AEs and SAEs | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>e</sup> | X | X | | X | | X | | | | | | | | X |
| Injection site reaction assessment <sup>f</sup> | | X | | X | X | X | X | X | X | X | X | X | X | X |
| Targeted physical examination | | | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>g</sup> | X | X | X | X | X | X | X | X | X | | | X | X | X |
| EFFICACY ASSESSMENTS | | | | | | | | | | | | | | |
| BILAG-2004 Index | X | X | | X | X | X | X | X | X | | | X | X | X |
| SLEDAI-2K | X | X | | X | X | X | X | X | X | | | X | X | X |
| PGA | X | X | | X | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | X | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | X | X | X | X | X | X | | | X | X | X |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |


Clinical Study Protocol: BOS161721-02

Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screena | Enroll | | | | Safe | ty Follo | w-Up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | - | | 10 | 11 | 12 |
| SLICC/ACR Damage Index | | X | | | | | | | X | | | | | |
| CCI | | X | | X | X | X | X | X | X | | | X | X | X |
| LABORATORY ASSESSMENT | ΓS | | | | | | | | | | | | | |
| CD4+ count | X | X | X | X | | X | | | X | | | | | |
| Clinical laboratory assessments (hematology and clinical | | | | | | | | | | | | | | |
| chemistry) <sup>h</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Coomb's test direct <sup>i</sup> | X | X | | X | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | X | X | | X | | | X | | | | | |
| Plasma CCI | X | X | | X | X | X | X | X | X | | | X | X | X |
| Plasma CCI & CCI | X | X | X | X | X | X | | | X | | | | | |
| Whole blood for leukocyte | | | | | | | | | | | | | | |
| immunophenotype | X | X | X | X | X | X | | | X | | | | | |
| ADA <sup>j</sup> | | X | X | X | X | X | | | X | | | | | X |
| nAb <sup>k</sup> | | | | | | X | | | X | | | | | |
| pSTAT3 <sup>1</sup> | | X | | X | X | X | | | X | | | | | |
| CCI | | X | | | | | | | X | | | | | |
| Whole blood RNA collection | | X | X | X | | X | | | | | | | | X |
| CCI | | | | | | | | | | | | | | |
| | X | X | | X | X | X | X | X | X | | | X <sup>m</sup> | X <sup>m</sup> | X <sup>m</sup> |
| CRP | X | | | | | X | | | | | | | | X |
| Serum pregnancy test (women) | X | | | | | | | | | | | | | |
| FSH (postmenopausal women) | X | | | | | | | | | | | | | |
| Urine pregnancy test (women) <sup>n</sup> | | X | | X | X | X | X | X | X | | | | | |
| TB test (QuantiFERON-TB Gold In-Tube) <sup>d</sup> | X | | | | | | | | | | | | | |
| Serology (hepatitis B and C,<br>HIV-1/2 combination) | X | | | | | | | | | | | | | |


Clinical Study Protocol: BOS161721-02

Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screena | Enroll | | | Tı | | Safe | ty Follo | w-Up | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 30 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 0 | $(\pm 3)$ | (± 3) | (±3) | (±3) | (±3) | (±3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | - | - | 10 | 11 | 12 |
| Stool sample <sup>o</sup> | X | | | | | | | | | | | | | |
| Spot urine for protein/creatinine | | | | | | | | | | | | | | |
| ratio | X | X | | X | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | X | X | X | X | X | X | | | X | X | X |
| PK Labs <sup>p</sup> | | | | | | | | | | | | | | |
| Predose <sup>q</sup> | | X | | X | X | X | X | X | X | | | | | |
| Postdose | | | X | | | | | | | X | X | X | X | X |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CC ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index; CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CC ; FSH = follicle stimulating hormone; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; RNA = ribonucleic acid; RNP = ribonucleoprotein; SAE = serious adverse event; SC = subcutaneous; CC ; SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; TDAR = T-cell dependent antigen response.

- <sup>a</sup> Screening assessments will be performed over more than 1 visit.
- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day). See Section 5.6.1 for further details.
- Randomization should occur after patient eligibility has been confirmed. The actual randomization procedure can be completed on Day -1 after eligibility confirmation or the morning of Day 0 prior to dosing for logistical purposes.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).
- <sup>c</sup> ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.
- Injection site reaction assessments to be performed predose and at 2 hours postdose.
- Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled outpatient days in the table above (excluding PK-only site visits at Days 187 and 195). When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.
- h Clinical laboratory assessments will include a fasting glucose and lipid panel, with exception of screening (Visit 1) which will be nonfasting.


Clinical Study Protocol: BOS161721-02

Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screena | Enroll | | | Tı | reatment | Period 1 | Follow-u | p | | | Safet | ty Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -28 | | 15 | 15 30 60 90 120 150 180 187 195 210 | | | | | | | | | | 270 |
| Days | to -1 | 0 | (± 3) | (± 3) | (±3) | (± 3) | (±3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | - | - | 10 | 11 | 12 |

When clinically indicated.


Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.

<sup>&</sup>lt;sup>k</sup> nAb is assessed if patient is positive for ADA.

Predose (trough) samples only.

only CCI collected during safety follow-up visits.

<sup>&</sup>lt;sup>n</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.

Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

PK samples will only be collected at the investigational sites that will be participating in the PK portion of the study.

<sup>&</sup>lt;sup>q</sup> Predose samples occur on study drug administration visit days.

#### 5 POPULATION

# 5.1 Participant Recruitment

Advertisements approved by the IRB, and investigator databases, may be used as recruitment procedures for adult men and women with moderately to severely active SLE.

#### **5.2** Number of Patients

Approximately 186 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD Phase 1b study, and approximately 156 patients will be randomized in the POC Phase 2 study. Note that approximately 30 dropouts are assumed.

# 5.3 Patient Screening

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Section 4.3]) for this study must be performed between Day -28 and Day -1.

#### 5.4 Inclusion Criteria

Patients who meet the following criteria will be considered eligible to participate in this clinical study:

- 1. Men and women, ages 18 to 70 years, inclusive
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion or Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory
  - c. C3 or C4 below normal as determined by central lab

- 5. At screening, the SLE Disease Activity Index 2000 (SLEDAI-2K) must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - ii. Points from lupus headache and organic brain syndrome will also be excluded
- 6. On Day 0, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - ii. Points from lupus headache and organic brain syndrome are also excluded
- 7. Patients must have at least 1 of the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - i. "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis in ≥ 2 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living that has been present on several days cumulatively over the past 4 weeks, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
      - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):
        - Ambulation, toileting, grooming- including bathing and dressing; feeding oneself, (and not responsive to steroids up to 10 mg/day, antimalarials, NSAIDs)
    - ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in ≥ 1 joint, (observed or throughout history), with some loss of functional range of movements which lead to some loss of functional range of motion as manifested by effects on instrumental ADLs such as:

- Cooking, driving, using the telephone or computer, shopping, cleaning, etc, and has been present on several days over the last 4 weeks, and is present at the time of the screening visit
- c. If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores
- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX)
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization) (see APPENDIX 3)
- 9. Women of childbearing potential (WOCBP; see Section 5.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  - b. Must not be breastfeeding
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

#### 5.5 Exclusion Criteria

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE)
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed
- 3. Any major surgery within 6 weeks of study drug administration, (Day 0), or any elective surgery planned during the course of the study
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB
  - b. History of active TB
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed.
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study. (See Section 5.6 for prohibited concomitant medication)
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic antibiotics or hospitalization
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
- 12. Cryptosporidium in the stool sample at screening
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening
- 15. CD4+ count < 500/µL at screening
- 16. Platelets < 50,000/mm $^3$  (50  $\times$  10 $^9$ /L) or < 35,000/ mm $^3$  (35  $\times$  10 $^9$ /L) if related to SLE, at screening
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if due to anemia related to SLE
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol)

19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockeroft-Gault calculation<sup>39</sup>:

GFR = ([1 for male] or [0.85 for female]) 
$$\times$$
 (140 – Age)  $\times$  BW / (72  $\times$  Creatinine)

- 20. Serum ALT and/or serum AST  $> 2 \times ULN$  at screening, unless explicitly related to lupus based on the investigator's judgment
- 21. Creatinine kinase (CK)  $> 3.0 \times$  ULN at screening, unless it is related to lupus myositis
- 22. Direct bilirubin  $> 1.5 \times ULN$  at screening (unless related to Gilbert's syndrome)
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (eg, IgG protein) or molecules made of components of monoclonal antibodies
- 25. History substance and/or alcohol abuse or dependence within the past 1 year, at the investigator's judgment
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision)
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4 or 5 on the Columbia Suicide severity Rating Scale (C-SSRS)
- 31. Current or pending incarceration
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness

#### **5.6** Concomitant Medications

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Patients should stay on stable regimen of other concomitant medications for the treatment of SLE (eg, analgesics, NSAIDs, statins, ACE

inhibitors/ARBs and other antihypertensive drugs), unless changes in these treatments are clinically indicated. Use of any other drugs for non-SLE conditions, including over-the-counter medications and herbal preparations, should remain stable unless change or addition is clinically necessary. Discussion with the medical monitor prior to initiation of new medication is strongly recommended. Any concomitant therapies must be recorded on the eCRF. Prior and concomitant medication use will be recorded for the 30 days prior to screening until the last follow-up visit. In addition, historical treatment for SLE (including immunosuppressant, anti-malarial, corticosteroid, and/or biologic agent) will be recorded for the 48 weeks prior to screening in the eCRF.

#### 5.6.1 Oral Corticosteroid Dose

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 0 (randomization day).

After Day 0 (after initiation of study therapy), no up-titration above 10 mg/day is allowed except for up to 1 CS burst for increased disease activity.

Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits.

- Once a patient has received the first dose of study drug, prednisone (or prednisone equivalent) may be tapered down at the discretion of the investigator
  - O Tapering is allowed after randomization except within 60 days of the primary (Day 210) and secondary (Day 120) endpoint assessments. Between Day 60 and Day 120, and between Day 150 and Day 210, oral CS doses must be held constant otherwise the patient will be declared a non-responder in efficacy assessments.

A maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed during the study between Day 0 and Day 60, according to the following:

- An oral CS "burst" between Day 0 and Day 60; (an increase of ≤ 40 mg/day of prednisone or equivalent), which must be tapered down to a maximum of 10 mg/day within 2 weeks of initiation of the "burst"
  - Alternatively, a single intramuscular (IM) dose of methylprednisolone (40 mg or equivalent) is permitted
  - o The course of the oral CS "burst" is not permitted to extend beyond Day 60

Treatment with inhalational CS therapy (eg, for asthma), or by any other route, is allowed. Other concomitant medications for SLE need to be taken at stable doses as per the inclusion criteria (Section 5.4).

#### **5.6.2** Other Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken prior to study drug administration and during the study are described below, and washout requirements are provided in APPENDIX 4. Medications taken within 30 days prior to screening must be recorded on the eCRF.

- 1. Prior exposure to BOS161721
- 2. Patients who have received treatment with anti-CD20 monoclonal antibodies within 6 months of screening; recovery of B cells (CD19+) must be documented (record absolute number of CD19+ B cells)
- 3. Patients who have received treatment with cyclophosphamide within the 1 year prior to screening
- 4. Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria (oral or topical) within 3 months of screening
- 5. Patients who are currently receiving or are scheduled to receive plasmapheresis or lymphapheresis therapy, or have received such therapy within 8 weeks prior to screening
- 6. Patients who have received any live vaccines within 30 days of screening. Note: Furthermore, live vaccines should not be used during the course of the study and within the 2 months following last dose. Other inactivated vaccines such as tetanus, etc, may be used according to local guidelines during treatment period
- 7. Patients who are scheduled or anticipated to have elective surgery during the course of the study
- 8. Initiation of new immunosuppressant or anti-malarial agent is not permitted. Note: Dose reduction or replacement may be allowed due to intolerability or shortage for patients on a stable dose prior to study initiation

# 5.7 Women of Childbearing Potential

WOCBP is defined as any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) and is not postmenopausal.

See Section 5.7.2 for detailed information regarding contraceptive requirements for WOCBP.

### **5.7.1 Determination of Menopause**

Menopause is defined as at least 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes. Women under the age of 55 years must have a documented serum FSH level > 40 mIU/mL at screening to confirm menopause.

### 5.7.2 Contraception

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion.

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion.

Investigators shall counsel WOCBP and men who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and men who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, patients must agree to the use of 1 method of highly effective contraception from the following:

- Male condoms with spermicide
- Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as 1 of the acceptable methods of contraception since they will not be receiving study drug.
- IUDs, such as ParaGard®
- Vasectomy
- Complete abstinence, defined as complete avoidance of heterosexual intercourse, is an
  acceptable form of contraception. Women who are abstinent while participating in the study
  must continue to have pregnancy tests. Acceptable alternate methods of highly effective
  contraception must be discussed in the event that the patient chooses to forego complete
  abstinence.

Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing.

### 5.8 Deviation from Inclusion/Exclusion Criteria

Deviation from the inclusion or exclusion criteria will not be allowed. If deviation of inclusion/exclusion criteria is discovered after randomization, the investigator should contact the medical monitor for discussion. A decision will be made whether to allow a patient continue or withdrawal from the study medication.

See Section 7.8 for additional details.

### 5.8.1 Patient Withdrawal and Replacement

See Section 6.5 for reasons for removal from the trial. Withdrawn patients may be replaced during the MAD study after discussion between the principal investigator or designee and sponsor.

#### 6 STUDY PROCEDURES

Refer to the eCRF completion guidelines for data collection requirements and documentation of study assessments/procedures.

# 6.1 Screening

Screening will be the same for both the MAD and POC studies.

Screening will take place from Day -28 to Day -1, and assessments may be performed over more than 1 visit. Confirmation that the most current IRB/IEC approved informed consent form (ICF) has been signed must occur before any study-specific screening procedures are performed. Procedures that are part of standard of care are not considered study-specific procedures and may be performed prior to informed consent and used to determine eligibility.

All screened patients will be assigned a unique screening number. The screening number will include a 3-digit site number and a 4-digit sequential number to identify patients from the time of screening. Only eligible patients who are confirmed by central review as meeting the inclusion/exclusion criteria, listed in Section 5.4 and Section 5.5 respectively, will be enrolled in the study. Screened patients who drop out of the clinical study before randomization will be recorded as screen failures. If rescreening occurs, the site will assign a new screening number.

Specific procedures at the screening visit will include:

- Medical history documentation
- Review of inclusion and exclusion criteria
  - o Patient medical records must contain documentation of SLE diagnosis
  - o C-SSRS
- Concomitant medication documentation
- Demographics
- Full physical examination
- Vital signs

- Chest x-ray
- Laboratory evaluations (nonfasting):
  - Hematology and clinical chemistry
  - o Serology (Hepatitis B and C; HIV-1/2 combination)
  - o TB test
  - o CRP
  - Direct Coomb's test (if indicated)
  - CD4+ count, total IgG and IgM levels, plasma CCI, plasma CCI, whole blood for leukocyte immunophenotype; CCI
  - Serum pregnancy test (WOCBP)
  - o FSH (postmenopausal women)
  - o Spot urine for protein/creatinine ratio
  - Urinalysis
  - Stool sample
- 12-lead ECG
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, Physician's Global Assessment (PGA) of disease activity

Screening procedures are listed in the Schedule of Assessments (Section 4.3), and details are provided in Section 7.

### 6.1.1 Retesting During Screening Period

A single retesting of laboratory parameters and/or other assessments during the screening period is permitted (in addition to any parameters that require a confirmatory value) only if:

- medically indicated
- there is evidence a laboratory sample was mislabeled, inadequately processed, and/or deteriorated in transit to the central laboratory

Any new result will override the previous result (ie, the most current result prior to randomization) and is the value by which study inclusion/exclusion will be assessed, as it

represents the patient's most current clinical state. This will also apply to patients who are being rescreened.

# 6.2 Enrollment/Randomization and Day 0 Treatment

Randomization should occur after patient eligibility for enrollment has been confirmed by the central eligibility review.

The study site will obtain a randomization number when registering the patient in IWRS. All patients will receive BOS161721 or placebo according to the kit number assigned by the IWRS randomization scheme.

After randomization, procedures include:

- PROs: CCI
- C-SSRS
- Laboratory evaluations (fasting):
  - Hematology and clinical chemistry
  - Direct Coomb's test (if indicated)
  - CD4+ count, total IgG and IgM levels, plasma CCl , plasma CCl , whole blood for leukocyte immunophenotype
  - o ADA
  - o pSTAT3 (predose [trough] samples only in Phase 2)
  - o CCI
  - Whole blood RNA collection
  - o CCI
  - See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies
  - o Urine pregnancy test will be collected on WOCBP prior to study drug administration
  - o Spot urine for protein/creatinine ratio
  - o Urinalysis
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 7.2.2.5 on SAE reporting requirements)

- Full physical examination
- Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours postdose on Day 0)
- 12-lead ECG (prior to PK blood draw)
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, PGA)
- SLICC/ACR damage index
- Study drug administration:
  - Administration of BOS161721 or placebo will take place on-site, and is discussed in Section 8.3
- Injection site reaction assessment, predose, and 2 hours postdose

Procedures on Day 0 are listed in the Schedule of Assessments (Section 4.3), and details are provided in Section 7.

All patients who are enrolled, randomized, and receive study drug, or undergo study-specific procedures should reconsent with any updated versions of IRB/IEC approved informed consents during study participation as applicable and per institutional guidelines.

# 6.3 Treatment Period/Follow-Up Visits

The following procedures will be performed as indicated in the Schedule of Assessments (Table 1 and Table 2). See Schedule of Assessment tables for allowable windows for each visit.

- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Concomitant medication documentation
- Documentation of AEs and SAEs (see Section 7.2.2.5 on SAE reporting requirements)
- PROs: CC
- Urine pregnancy tests will be collected on WOCBP prior to study drug administration
- Injection site reaction assessments will be performed predose and 2 hours postdose
- Direct Coomb's test (if indicated)
- Spot urine for protein to creatinine ratio
- Urinalysis

- CCI
- Plasma CCI
- PGA, BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, and the CLASI will be completed
- SLICC/ACR Damage Index will be completed at Day 180
- C-SSRS
- ECGs prior to PK blood draw
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies, respectively
- Fasting hematology and chemistry assessments
- The CD4+ count and total IgG and IgM levels
- Plasma CC & CC , ADA, and whole blood for leukocyte immunophenotype
- pSTAT3
- Whole blood RNA
- CRP and nAb will be assessed if patient is positive for ADA
- CCI

### 6.4 Safety Follow-Up Visits

Safety follow-up visits will take place at Days 210, 240, and 270. These visits will include the following assessments as indicated in the Schedule of Assessments (Table 1 and Table 2):

- PROs: CC
- Documentation of AEs and SAEs (see Section 7.2.2.5 on SAE reporting requirements)
- Injection site reactions
- Targeted physical examination
- Vital signs (prior to PK blood draw)
- Spot urine for protein/creatinine ratio and urinalysis
- Concomitant medication documentation

- BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, and PGA
- Fasting clinical laboratory assessments (hematology and clinical chemistry)
- Direct Coomb's test (if indicated)
- Plasma CCI
- CCI
- pSTAT3
- 12-lead ECG (prior to PK blood draw)
- CRP
- ADA
- Whole blood RNA collection
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies, respectively

#### 6.5 Premature Discontinuation

While patients are encouraged to complete all study evaluations, they may withdraw from the study at any time and for any reason. Every effort will be made to determine why any patient withdraws from the study prematurely. If the patient is unreachable by telephone, a registered letter, at the minimum, should be sent to the patient requesting him/her to contact the clinic.

All patients who withdraw from the study with an ongoing AE or SAE must be followed until the end of study or until the event is resolved or deemed stable, respectively.

If a patient withdraws prematurely after dosing, an end of treatment (EOT) visit should be performed (Day 180) and a last follow-up visit 90 days after dosing should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 6.4).

Patient participation may be terminated prior to completing the study and the reason recorded as follows:

- AE/SAE
- Protocol deviation
- Lost to follow-up
- Patient withdraws consent at their own request

- Investigator decision
- Decision by sponsor (other than AE/SAE, protocol deviation, or lost to follow-up)

Withdrawn patients may be replaced after discussion between the investigator or designee and sponsor.

#### 7 ASSESSMENTS

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances, outside of the control of the investigator, which may make it unfeasible to perform the test. In these cases, the investigator will take all steps necessary to ensure the safety and wellbeing of the patient. When a protocol required test cannot be performed the investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. All protocol violations are entered directly into the eCRFs.

### 7.1 Medical History, Demographic and Other Baseline Information

The medical history comprises:

- General medical history
- Documentation of SLE diagnosis
- Historical medication therapy for SLE

The following demographic information will be recorded:

- Age
- Ethnic origin (Hispanic/Latino or not Hispanic/not Latino)
- Race (White, American Indian/Alaska Native, Asian, Native Hawaiian or other Pacific Islander, Black/African American)
- Height (without shoes, in cm)
- Body weight, without shoes (kg)
- Body mass index (BMI [kg/m<sup>2</sup>])

Other baseline characteristics will be recorded as follows:

- Concomitant medication documentation (see Section 5.6)
- Status of child bearing potential and contraception

# 7.2 Safety Assessments

# 7.2.1 Laboratory Assessments

Laboratory tests will be performed at times defined in the Schedule of Assessments (Section 4.3). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

A central laboratory will be used (with the exception of urine pregnancy tests and stool analysis) to ensure accuracy and consistency in test results. The central laboratory will transmit all results for protocol tests, scheduled and unscheduled, to the clinical data base. Laboratory/analyte results that could unblind the study (ie, biomarker results) will not be reported to investigative sites. Urinalysis will be performed on midstream, clean catch specimens. Some biomarkers listed above will not be drawn at some sites due to geographical logistical challenges. See the laboratory manual for details.

Endpoint analyses will be based on changes from baseline assessments at Days 120 and 210.

Table 3. Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| Hemoglobin | BUN | рН | Spot urine for protein/creatinine ratio |
| Hematocrit | Creatinine | Glucose (qual) | FSH <sup>b</sup> |
| RBC count | Glucose (fasting) | Protein (qual) | Urine pregnancy test <sup>c</sup> |
| RDW | Calcium | Blood (qual) | QuantiFERON®-TB Gold In-Tube test |
| MCV | Sodium | Ketones | (QFT-G) |
| MCH | Potassium | Nitrites | Serology <sup>d</sup> (Hepatitis B and C; HIV-1/2 |
| MCHC | Chloride | Leukocyte esterase | combination) |
| Platelet count | Total CO <sub>2</sub> (bicarbonate) | Urobilinogen | Stool sample <sup>e</sup> |
| WBC count | AST, ALT | Urine bilirubin | |
| CD4+ count | Total bilirubin | Microscopy <sup>a</sup> | |
| Total neutrophils (Abs) | Alkaline phosphatase | | |
| Eosinophils (Abs) | Creatine kinase | | |
| Monocytes (Abs) | Uric acid | | |
| Basophils (Abs) | Albumin | | |
| Lymphocytes (Abs) | Total cholesterol | | |
| Reticulocytes (%) | (fasting) | | |
| | LDL-C (fasting) | | |
| | HDL-C (fasting) | | |
| | Triglycerides (fasting) | | |
| | Total protein | | |
| | PT/INR | | |
| | Additional Tests <sup>f</sup> | | Immunogenicity, PD and other<br>Biomarker Tests |
| | (potential Hy's Law) | | |
| | AST, ALT (repeat) | | ADA |
| | Total bilirubin (repeat) | | nAb <sup>g</sup> |
| | Albumin (repeat) | | pSTAT3 (predose [trough] samples |
| | Alkaline phosphatase | | only, in Phase 2) Total IgG & IgM |
| | (repeat) Direct bilirubin | | Plasma CCI |
| | Indirect bilirubin | | Plasma CCI & CCI |
| | GGT | | Whole blood for leukocyte |
| | UUI | | immunophenotype and RNA |
| | | | CC |
| | | | CCI |
| | | | Antibodies CC |
| | | | CRP |

Abbreviations: Abs = absolute; ADA = anti-drug antibody; ALT = alanine aminotransferase;

; AST = aspartate aminotransferase; BUN = blood urea

Direct Coomb's testh

nitrogen; C = complement; CD4+ = cluster of differentiation 4; CRP = C-reactive protein;

dsDNA = double-stranded deoxyribonucleic acid;; FSH = follicle stimulating hormone;

GGT = gamma-glutamyltransferase; HDL-C = high-density lipoprotein cholesterol; HIV = human

immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; INR = international normalized ration; IL-21 = interleukin 21; LDL-C = low-density lipoprotein cholesterol; MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = Mean corpuscular volume; nAb = neutralizing antibody; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; PT = prothrombin time; qual = qualitative; RBC = red blood cell; RDW = RBC distribution width; RNA = ribonucleic acid;

**Table 3.** Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| RNP = ribonucleopr | otein; SAE = serious advers | se event; SC = subcutane | ous; CCI |
| CCI | ; $TB = tuber$ | culosis. | |

- a. On all urine samples.
- b. At screening only, in women who are amenorrheic for at least 12 consecutive months and under 55 years old.
- c. For WOCBP.
- d. Screening only.
- At screening, and if a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- f. Additional testing for potential Hy's Law cases only (See Section 7.2.2.6.3).
- g. If patient is positive for ADA.
- If clinically indicated.

#### 7.2.1.1 Pregnancy testing

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits prior to study drug administration, and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be discontinued from study drug, an EOT visit should be performed (Day 180), and a last follow-up visit 90 days after last dose should be scheduled (Day 270). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 6.4).

See Section 7.2.2.7.1 for information on reporting of pregnancies as AEs/SAEs during the study.

### 7.2.1.2 Tuberculosis Screening

During the screening period, it must be determined and documented that a patient does not have evidence of active or latent or inadequately treated TB per the exclusion criteria (Section 5.5). The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 0).

# 7.2.1.2.1 Mycobacterium Tuberculosis Testing Using QuantiFERON Test<sup>40</sup>

QuantiFERON®-TB Gold In-Tube (QFT-G) is an in vitro diagnostic test using a peptide cocktail simulating ESAT-6, CFP-10, and TB 7.7 proteins to stimulate cells in heparinized whole blood. Detection of INFγ performed by enzyme-linked immunosorbent assay (ELISA) is used to identify in vitro responses to these peptide antigens that are associated with Mycobacterium tuberculosis infection. QFT-G is an indirect test for M. tuberculosis infection (including disease) and is intended for use in conjunction with risk assessment, radiography and other medical and diagnostic evaluations.

Test results will be reported as positive, negative, or indeterminate. A negative QFT-G test result is required to meet the inclusion criterion. In the case of an indeterminate result, repeat tests should be permitted for the purpose of determining eligibility of patients to enroll in this study. If a repeat test is indeterminate again, the patient is a screen failure. The procedure for using this test and interpreting the results will be described fully in the laboratory manual, which will be provided to investigators.

#### 7.2.2 Adverse Events

#### 7.2.2.1 Definitions

An AE is defined as any untoward medical occurrence experienced by a study patient, whether or not considered drug related by the principal investigator.

AEs are unfavorable changes in a general condition, subjective or objective signs or symptoms, worsening of pre-existing concomitant disease, and clinically significant abnormality in laboratory parameters observed in a patient in the course of a clinical study.

Non-serious SLE manifestations or abnormal laboratory results related to SLE disease activity would not be recorded as AEs unless they meet the definition for SAEs (Section 7.2.2.5).

# 7.2.2.2 Recording of Adverse Events

AEs should be collected and recorded for each patient from the date of the first dose of study drug until the end of their participation in the study, including the safety follow up period.

AEs may be volunteered spontaneously by the study patient, or discovered by the study staff during physical examinations or by asking an open, nonleading question such as 'How have you been feeling since you were last asked?' All AEs and any required remedial action will be recorded on the Adverse Events eCRF and Safety Adverse Event Form. The details of the AE, date of AE onset (and time, if known), date of AE outcome (and time, if known), and action taken for the AE will be documented together with the principal investigator's assessment of the seriousness of the AE and causal relationship to the study drug and/or the study procedure.

All AEs should be recorded individually, using diagnostic terms where possible. If the diagnosis is not established, individual symptoms may be reported. The AEs will subsequently be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

#### **7.2.2.3** Severity of Adverse Events

Each AE will be assessed by the principal investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 criteria. <sup>41</sup> When changes in the severity (grade) of an AE occur more frequently than once a day, the maximum severity for the event should be noted for that day. Any change in severity of signs and symptoms over a number of days will be captured by recording a new AE, with the amended severity grade and the date (and time, if known) of the change.

### 7.2.2.4 Causality of Adverse Events

The principal investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (Table 4) should be selected based on medical judgment, considering the definitions below and all contributing factors.

| Table 4. | Causality Definitions |
|---|---|
| Related | A clinical event, including laboratory test abnormality, occurs in a plausible time relationship to treatment administration and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (dechallenge <sup>a</sup> ) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge <sup>b</sup> procedure if necessary. |
| Unrelated | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative dechallenge and rechallenge information. Typically explained by extraneous factors (eg, concomitant disease, environmental factors, or other drugs or chemicals). |

Dechallenge: Upon discontinuation of a drug suspected of causing an AE, the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation (positive dechallenge), or the symptoms continue despite withdrawal of the drug (negative dechallenge). Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia).

Rechallenge: Upon re-administration of a drug suspected of causing an AE in a specific patient in the past, the AE recurs upon exposure (positive rechallenge), or the AE does not recur (negative rechallenge).

An unexpected adverse drug event is any adverse drug event for which the specificity or severity is not consistent with the current IP.

#### 7.2.2.5 Seriousness of Adverse Events

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life threatening; this means that the patient was at risk of death at the time of the event; it does not mean that the event hypothetically might have caused death if it were more severe
- Requires hospitalization or prolongation in existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly or birth defect
- Is another important medical event (see below)

Important medical events that do not result in death, are not life threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such events are:

- Intensive treatment in an emergency room or at home for allergic bronchospasm
- Blood dyscrasias or convulsions that do not result in inpatient hospitalization
- Development of drug dependency or drug abuse

Hospitalization for elective surgery or routine clinical procedures that are not the result of AE (eg, elective surgery for a pre-existing condition that has not worsened) need not be considered SAEs. If anything untoward is reported during the procedure, that occurrence must be reported as an AE, either 'serious' or 'nonserious' according to the usual criteria.

Suspected unexpected serious adverse reactions (SUSARs) are AEs that are associated with the use of the drug and are serious and unexpected.

# **7.2.2.6** Adverse Events of Special Interest

AEs of special interest in this study include the following:

- 1. Anaphylaxis and serious allergic reactions
- 2. Injection site reaction, including erythema, pain, and induration
- 3. Drug Induced Liver Injury (DILI) assessed following Hy's Law
- 4. Malignancy
- 5. Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, and disseminated tuberculosis
- 6. Cryptosporidiasis

#### 7.2.2.6.1 Anaphylaxis and Serious Allergic Reactions

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria. <sup>42</sup> In the event of anaphylactic reaction or severe/serious hypersensitivity/allergic reaction, the patient must discontinue IP and emergency resuscitation measures implemented. In case of other mild to moderate hypersensitivity reaction, depending on the severity, the investigator may manage in accordance with the standard-of-care.

Anaphylaxis is highly likely when any one of the following 3 criteria is fulfilled:

1. Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (eg, generalized hives, pruritus, or flushing, swollen lips-tongue-uvula) and at least 1 of the following:

- a. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow [PEF], hypoxemia)
- b. Reduced blood pressure or associated symptoms of end-organ dysfunction (eg, hypotonia [collapse], syncope, incontinence)
- 2. Two or more of the following that occur rapidly after exposure to a likely allergen for that patient (minutes to several hours):
  - a. Involvement of the skin-mucosal tissue (eg, generalized hives, itch-flush, swollen lips-tongue-uvula)
  - b. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)
  - c. Reduced blood pressure or associated symptoms (eg, hypotonia [collapse], syncope, incontinence)
  - d. Persistent gastrointestinal symptoms (eg, crampy abdominal pain, vomiting)
- 3. Reduced blood pressure after exposure to known allergen for that patient (minutes to several hours):
  - a. Systolic blood pressure of less than 90 mm Hg or greater than 30% decrease from the patient's baseline

### 7.2.2.6.2 Injection Site Reactions

Injection site reactions are to be captured and reported as AEs. These may include injection site erythema, pain, and induration. The investigator should provide a clear description of the observed or reported AE including location and severity. All concomitant treatments used to treat injection site reactions should be recorded and captured in the eCRF, together with the AE of injection site reactions.

### 7.2.2.6.3 Potential Drug-Induced Liver Injury

Abnormal values in AST and/or ALT levels concurrent with abnormal elevations in total bilirubin level that meet the criteria outlined below in the absence of other causes of liver injury are considered potential cases of DILI, and as potential Hy's Law cases, and should always be considered important medical events. If symptoms compatible with DILI precede knowledge of serum chemical test abnormalities, liver enzyme measurements should be made immediately, regardless of when the next visit or monitoring interval is scheduled. In some cases, symptoms may be an early sign of injury and although typically less sensitive than serum enzyme elevations, they may indicate a need for prompt serum testing. An increase in liver enzymes should be confirmed by a repeated test within 48 to 72 hours following the initial test, prior to reporting of a potential DILI event. Patients will continue to have weekly or biweekly liver enzyme measurements until resolution or levels return to baseline.

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 7.2.2.7.2 for reporting details).

#### Potential DILI is defined as:

1. ALT or AST elevation  $> 3 \times ULN$ 

#### **AND**

2. Total bilirubin > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)

#### **AND**

3. No other immediately apparent possible causes of ALT or AST elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic

The patient should return to the investigational site and be evaluated as soon as possible, include laboratory tests, detailed history, and physical assessment. In addition to repeating measurements of AST and ALT, laboratory tests should include albumin, CK, total bilirubin, direct and indirect bilirubin, GGT, prothrombin time (PT)/International Normalized Ratio (INR), and alkaline phosphatase. A detailed history, including relevant information, such as review of ethanol, acetaminophen, recreational drug and supplement consumption, family history, occupational exposure, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and work exposure, should be collected. Further testing for acute hepatitis A, B, or C infection and liver imaging (eg, biliary tract) may be warranted. All cases confirmed on repeat testing as meeting the laboratory criteria defined above, with no other cause for liver function test (LFT) abnormalities identified at the time should be considered potential Hy's Law cases irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal LFTs. Such potential Hy's Law cases should be reported as SAEs.

Study drug discontinuation is considered if there is marked serum AST or ALT elevation or evidence of functional impairment (as indicated by rising bilirubin or INR, which represent substantial liver injury) that is related to study drug. Discontinuation of treatment should be considered if:

- ALT or AST > 8 × ULN
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks

Discontinuation of treatment must occur if:

- ALT or AST >3 × ULN and (total bilirubin > 2 × ULN or INR > 1.5)
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)

### 7.2.2.6.4 *Malignancy*

The identification of a malignancy event will be made by the study site and communicated to the sponsor or designee. AEs should be reported as serious per the criteria in Section 7.2.2.5.

After the first dose of study drug, when there is a decision to biopsy a potentially malignant tumor, lymph node, or other tissue, the investigator and/or consultant(s) should contact the sponsor clinicians or designee to discuss the issue and any decisions as soon as possible.

### 7.2.2.6.5 Specific Infections

Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, shingles, disseminated herpes simplex, or disseminated tuberculosis will be recorded as AEs of special interest.

Cryptosporidiosis is also considered an AE of special interest. Patients will be evaluated for cryptosporidium in the stool at screening, and as clinically indicated (eg, watery diarrhea) during the study. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

# 7.2.2.7 Reporting of Adverse Events

AE reporting will be carried out in accordance with applicable local regulations, including regulatory agency and IRB reporting requirements.

Each AE is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 7.2.2.7.2.

### 7.2.2.7.1 Reporting of Pregnancy

As information is available, a pregnancy diagnosed during the study will be reported within 24 hours to the sponsor via the Pregnancy Notification and Outcome Form, including pregnancy in female patients who received study drug and female partners of male study patients who received study drug. The pregnancy should be followed to term and/or outcome and this outcome should also be reported to the sponsor via the Pregnancy Notification and Outcome Form. Pregnancy itself is not regarded as an AE or SAE unless there is complication.

In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an AE or SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live born, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as serious adverse events when the investigator assesses the neonatal death as related or possibly related to exposure to investigational product.

# 7.2.2.7.2 Reporting of Serious Adverse Events

The principal investigator is responsible for providing notification to the sponsor of any SAE via the Safety Adverse Event Form, whether deemed study drug related or not, that a patient experiences during their participation in this study within 24 hours of becoming aware of the event.

If an SAE is fatal or life threatening, notification to the sponsor must be made aware immediately, irrespective of the extent of available AE information. This timeframe also applies to additional new information (follow-up) on previously forwarded SAE reports as well as to the initial and follow-up reporting of exposure during pregnancy and exposure via breastfeeding cases. In the rare event that the investigator does not become aware of the occurrence of an SAE immediately (eg, if an outpatient study patient initially seeks treatment elsewhere), the investigator is to report the event within 24 hours after learning of it and document the time of his/her first awareness of the AE.

The principal investigator will review each SAE and evaluate the intensity and the causal relationship of the event to the study drug. All SAEs will be recorded from the time of first dose of study drug through the safety follow-up period (up to Day 270). SAEs occurring after the final follow-up visit and coming to the attention of the principal investigator must be reported only if there is (in the opinion of the principal investigator) reasonable causal relationship with the study drug.

As a minimum requirement, the initial notification should provide the following information:

- Study number
- Patient number
- Details of the SAE (verbatim details are sufficient for immediate notification)
- Criterion for classification as 'serious'
- Causality assessment (which may be updated in a follow-up report when sufficient information is available to make this classification)

Initial reports of SAEs must be followed later with detailed descriptions, including clear photocopies of other documents as necessary (eg, hospital reports, consultant reports, autopsy reports, etc), with the study patient's personal identifiers removed. All relevant information

obtained by the principal investigator through review of these documents will be recorded and submitted to the sponsor within 24 hours of receipt of the information. If a new Safety Adverse Event Form is submitted, then the principal investigator must sign and date the form. The sponsor may also request additional information on the SAE, or clarification of omitted or discrepant information from the initial notification, which the principal investigator or an authorized delegate should submit to the sponsor within 24 hours of the request as possible.

### 7.2.2.7.3 Reporting of Adverse Events of Special Interest

AEs of special interest will be reported to safety immediately or within 24 hours of the site becomes aware of the event and recorded as such on the Adverse Events eCRF and Safety Adverse Event Form.

Potential DILI will be reported based on specifications mentioned in Section 7.2.2.6.3.

Each AE of special interest is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 7.2.2.7.2.

### **7.2.2.8** Follow Up of Adverse Events

All AEs will be followed up through the safety follow-up visits. All SAEs experienced by a patient, irrespective of the suspected causality, will be monitored until the event has resolved, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the principal investigator and medical monitor, until there is a satisfactory explanation for the changes observed, or until the patient is lost to follow-up.

See Section 7.2.2.7.1 for details related to follow-up of pregnancy. See Section 7.2.2.6.3 for details related to follow-up of potential DILI. See Section 7.2.2.6.4 for details related to follow-up of malignancy.

#### 7.2.3 Vital Signs

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (Section 4.3). Vital signs will be assessed on Day 0 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study (excluding PK-only site visits). Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq 5$  minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

### 7.2.4 12-Lead Electrocardiograms

ECG will be assessed as specified in the Schedule of Assessments (Section 4.3). ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

The ECG will include all 12 standard leads and a Lead II rhythm strip on the bottom of the tracing. The ECG will be recorded at a paper speed of 25 mm/second. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QT interval corrected for heart rate using Fridericia's formula (QTcF).

All ECGs must be evaluated by a qualified physician or qualified designee for the presence of abnormalities and will be captured electronically and retained for future evaluation if required, up to the time of the clinical study report (CSR) completion.

### 7.2.5 Physical Examinations

The full physical examination will be completed at screening and Day 0. It includes an assessment of general appearance and evaluation of head, eyes, ears, nose, mouth, throat, neck, thyroid, lymph nodes, and extremities, and dermatologic, respiratory, cardiovascular, gastrointestinal, musculoskeletal, neurologic, and psychiatric systems.

The targeted (limited) physical examination will be completed at all other visits as indicated in the Schedule of Assessments (Section 4.3). It includes evaluation of patient complaints and SLE disease-related issues, and will exclude the genitourinary system.

#### 7.2.6 C-SSRS

The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed by Columbia University researchers for the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening. 43

The C-SSRS evaluation will be performed as specified in the Schedule of Assessments (Section 4.3). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

### 7.2.7 Injection Site Reactions

Patients will be monitored for local injection site reactions as specified in the Schedule of Assessments (Section 4.3). Local injection site reactions will be assessed predose and at 2 hours postdose. Injection site reactions should be managed according to the standard of care. Injection site reactions are to be reported as AEs of special interest (see Section 7.2.2.7.3).

#### 7.2.8 Immunogenicity

The serum samples to measure the presence of ADA will be collected as specified in the Schedule of Assessments (Section 4.3). Blood samples (4 mL) to provide approximately 1.5 mL

of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K<sub>2</sub>EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.

After the first dose, if a patient tests positive in the validated confirmatory ADA assay, the sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay.

# 7.3 Efficacy Assessments

All efficacy assessments will be performed at times defined in the Schedule of Assessments (Section 4.3).

#### **7.3.1 SLEDAI-2K**

The SLEDAI-2K is a validated instrument that measures disease activity in SLE patients at the time of the visit and in the previous 30 days. It is a global index and includes 24 clinical and laboratory variables that are weighted by the type of manifestation, but not by severity. The total score falls between 0 and 105, with higher scores representing increased disease activity. The SLEDAI-2K has been shown to be a valid and reliable disease activity measure in multiple patient groups. A SLEDAI -2K of 6 or more generally represents moderately to severely active disease. 44

#### 7.3.2 BILAG 2004

The BILAG-2004 index is an organ-specific 97-question assessment based on the principle of the doctor's intent to treat. Only clinical features attributable to SLE disease activity are to be recorded and based on the patient's condition in the last 4 weeks compared with the previous 4 weeks. It will be scored as not present (0), improved (1), the same (2), worse (3), or new (4). Disease activity is graded separately for 9 body systems to 5 different grades (A to E) as follows: A ("Active") is very active disease, B ("Beware") is moderate activity, C ("Contentment") is mild stable disease, D ("Discount") is inactive now but previously active, and E ("Excluded") indicates the organ was never involved. A shift from BILAG-2004 Grade A or B to a lower grade indicates a clinically relevant change in disease activity as the BILAG-2004 grades mirror the decision points for treatment interventions.

Only investigators that complete BILAG-2004 training will be allowed to perform the BILAG-2004 assessments. Preferably, the same investigator should evaluate the patient at each BILAG-2004 assessment from screening to study completion. The investigator must maintain documentation with descriptive details supporting the BILAG-2004 scoring (eg, chart, worksheet, clinic notes, and labs) at each visit.

See APPENDIX 5 for detailed specifications.

### 7.3.3 PGA of Disease Activity

The PGA is used to assess investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients".

When scoring the PGA, the assessor should always look back at the score from the previous visit.

### 7.3.4 Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response

### **7.3.4.1 SRI-4 Response**

Patients will be evaluated for SRI-4 scores at Day 210, with evaluation for sustained reduction of oral CS (< 10 mg/day and < Day 0 dose) between Day 120 and Day 210.

The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. Response based on the SRI-4 is defined by:

1)  $\geq$  4-point reduction in SLEDAI-2K global score, 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B), and 3) no deterioration from baseline in the PGA by  $\geq$  0.3 points. The SRI-4 response in patients with moderate to severe SLE is associated with broad improvements in clinical and patient-reported outcomes. <sup>45</sup>

Each patient, after providing their Day 210 visit SRI-4 response, will be evaluated as either a responder or non-responder.

### 7.3.4.2 SRI-5 and SRI-6 Response

Like the SRI-4, the SRI-5 and SRI-6 are composite indices of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. However, the SRI-5 and SRI-6 are computed with a minimal three-point or five-point improvement in SLEDAI-2K being required, respectively. 46

The SRI-5 and SRI-6 are evaluated for response at Day 180, along with a sustained reduction of oral CS ( $\leq$  10 mg/day and  $\leq$  Day 0 dose) between Day 120 and Day 210.

#### 7.3.4.3 BICLA Response

The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and PGA. BICLA response is defined as 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (eg, all B [moderate disease] scores falling to C [mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4)  $\leq$  10% deterioration in PGA score and 5) no treatment failure. 44 It is driven primarily by the BILAG, and has been used in Phase 2 and 3 mAb studies. 47

For the endpoints of BICLA response at Days 210, 240, and 270, patient scores will be completed and response determined.

### 7.3.5 CLASI Response

The CLASI is a comprehensive tool for assessment of disease activity and damage in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity. <sup>48</sup> Response is defined as 50% improvement from baseline in "A" or "B" scores. This assessment will be applied to all patients as all are required to have cutaneous disease activity.

For the secondary efficacy endpoint of CLASI response at Day 210, patient scores on MAD and POC studies will be compared with baseline for 50% improvement.

#### 7.3.6 ACR-28 Joint Count

The ACR-28 joint count will evaluate the number of tender and swollen joints in the shoulder, elbow, wrist, hand, knee joints. Joints of the feet are excluded.

#### 7.4 Other Variables

### 7.4.1 SLICC/ACR Damage Index

The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in patients with SLE regardless of cause, with demonstrated content, face, criterion, and discriminant validity. It will be performed on Days 0 and 180.

#### 7.4.2 **PROs**

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the CCI and the CCI and will be assessed as specified in the Schedule of Assessments (Section 4.3).




#### 7.5 Pharmacokinetic Assessments

During the MAD Phase 1b (all sites) and POC Phase 2 (select sites only) studies, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to Table 1 and Table 2.

PK parameters include the following:

•  $C_{max}$ ,  $T_{max}$ , AUC,  $t_{1/2}$ , CL,  $V_d$ 

Plasma concentrations of BOS161721 will be measured using a validated immunoassay. The PK parameters will be calculated from the plasma concentration-nominal time profiles for the IA2 and actual time profiles for the final analysis. The non-compartmental analysis will be performed using appropriately validated PK/PD software.

# 7.6 Pharmacodynamic Assessments

Blood samples for PD parameters (plasma) will be collected at times indicated in the Schedule of Assessments (Section 4.3) for each of the following parameters:

- pSTAT3
- Antibodies: CCl
- Plasma complement (CCI)
- Plasma CCI and CCI
- Whole blood for leukocyte immunophenotype
- Whole blood RNA
- IgG and IgM and CD4+ count

### 7.7 Pharmacokinetic/Pharmacodynamic Relationship

Evidence of any PK/PD relationships will be evaluated between BOS161721 plasma concentrations and the available PD endpoints and biomarkers.

### 7.8 Protocol Deviations

Protocol deviations will be documented during the study. Per the statistical analysis plan (SAP), these will be listed by patient and summarized by deviation category by treatment group.

### 8 STUDY DRUG MANAGEMENT

# 8.1 Description

#### 8.1.1 Formulation



Additional information regarding dose preparation will be provided in a separate Pharmacy Manual.

#### 8.1.2 Storage

All supplies of BOS161721 or placebo must be stored in accordance with the manufacturer's instructions. BOS161721 or placebo will be stored in a securely locked area, accessible to authorized persons only, until needed for dosing.

Information regarding storage and dose preparation will be provided in a separate Pharmacy Manual.

# 8.2 Packaging and Shipment

Investigational medicinal products will be supplied by Boston Pharmaceuticals, Inc. Investigational medicinal products will be packaged and labeled according to applicable local and regulatory requirements.

### 8.3 Dose and Administration

Details of dosing are provided in Section 4.1.

Each unit dose will be prepared by a qualified staff member. The vials of investigational product (IP) will appear identical and will have a "blinded" label on the vials that will state mg or placebo. When the site goes into the IWRS to request the patient kit(s), the IWRS will assign the appropriate number of kits (regardless of assignment to placebo or active treatment) per the dose (ie, CC).

If a patient is randomized to the placebo arm, they will receive the matching number of kits.

The designated staff member (or designee under the direction of the designated staff member) will dispense BOS161721 or placebo for each patient according to the protocol, randomization list, and Pharmacy Manual, if applicable.

After receiving sponsor approval in writing, the investigational site is responsible for returning all unused or partially used BOS161721 or placebo to the sponsor or designated third party or for preparing BOS161721 or placebo for destruction via incineration.

Further details are found in a separate Pharmacy Manual.

### 8.4 Accountability

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Products returned to the pharmacy will be stored under the same conditions as products not yet dispensed. The returned products should be marked as 'returned' and kept separate from the products not yet dispensed.

All dispensing and accountability records will be available for sponsor review after database lock procedures are completed. During safety monitoring, the drug accountability log will be reconciled with the products stored in the pharmacy.

# 8.5 Prohibited Concomitant Therapy

Prohibited concomitant medications are discussed in Section 5.6 and APPENDIX 4 and will be listed as protocol violations if taken when not permitted.

# 8.6 Compliance

Dosing will be performed by trained, qualified personnel designated by the principal investigator. The date and time of dosing will be documented on each dosing day. Comments will be recorded if there are any deviations from the planned dosing procedures.

### 9 STATISTICS

There are 2 IAs planned for the study. The first IA will be conducted at the time of the POC decision for dose selection. The second IA will be performed for futility (see Section 9.3). Before the first IA, a SAP will be finalized, providing detailed methods for the analyses outlined below. Any deviations from the planned analyses will be described and justified in the final integrated CSR.

The following standards will be applied for the analysis unless otherwise specified. Continuous data will be summarized by treatment group using descriptive statistics (number, mean, standard deviation [SD], minimum, median, and maximum). Categorical data will be summarized by treatment group using frequency tables (number and percentage).

# 9.1 Sample Size

Sample size in the Phase 1b study is based on operational consideration.

A summary of the power in the trial for the chosen sample size is provided in Table 5, with N = 132 randomized 89:43 to the chosen dose for the POC study and placebo, respectively; this includes 12 patients from the MAD study who were in the cohort of the mid or high dose if chosen for the POC study.

| Table 5. | Sample Siz | e |
|-----------|---------------|---|
| I WOIC CI | Swill pie Siz | • |

| Type 1 Error | TRUE Underlying<br>Response Rate (%) | | | Minimum OBSERVED Respons<br>Rates Yielding Statistical<br>Significance | |
|---|---|---|---|---|---|
| (1-Sided) | Placebo | Treatment | Overall Power | Placebo | Treatment |
| | 40 | 60 | 0.54 | | |
| 0.025 | 40 | 65 | 0.75 | 40 | 60 |
| | 40 | 70 | 0.9 | | |
| | 40 | 60 | 0.63 | | |
| 0.05 | 40 | 65 | 0.81 | 40 | 58 |
| | 40 | 70 | 0.93 | | |

Total sample size of approximately 156 patients is planned for analysis, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Note that approximately 36 dropouts are assumed.

### 9.2 Statistical Methods

### 9.2.1 Analysis Populations

The primary efficacy analysis will be based on the full analysis set (FAS), defined to be all patients with at least 1 baseline and post-baseline efficacy evaluation. A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be identified based on blinded data prior to unblinding the final analysis dataset. Safety analyses will be based on all patients who receive test treatment. Pharmacokinetic analysis will be conducted on the PK analysis set (PK), defined as the FAS with sufficient concentration data for the calculation of PK parameters. All analyses will combine data from the MAD and POC studies and focus on the active treatment dose chosen for the POC study versus placebo. The 0.05 1-sided type 1 error level is included for POC, and the 0.025 1-sided type 1 error level for potential use of this trial to support regulatory filing.

### 9.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized via appropriate summary statistics by treatment group and overall, for each phase of the trial.

# 9.2.3 Primary Endpoint(s)

The proportion of patients who achieve treatment response (measured by SRI-4 at Day 210 along with a sustained reduction of oral CS) will be analyzed via Cochran-Mantel-Haenszel (CMH) analysis. The primary endpoint will be analyzed on the FAS and if needed the PP analysis set. In addition, missing values will be addressed by employing a last observation carried forward (LOCF) analysis and/or other appropriate analytic approaches as a sensitivity analysis. Details will be available in the SAP.

### 9.2.4 Secondary Endpoint(s)

Binary efficacy endpoints will be assessed via CMH analysis. Continuous efficacy endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-by-time interaction, baseline covariate, and covariate-by-time interaction. The secondary efficacy endpoint will be analyzed on the FAS and if needed the PP analysis set. Details will be available in the SAP.

### 9.2.5 Analysis of Safety

### 9.2.5.1 Safety Analysis

Safety analyses will be performed on the Safety Analysis Set. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. Incidences (number and percent) of AEs will be presented by treatment group. Incidences of AEs will also be presented by maximum severity and relationship to study medication. For the MAD study, the placebo patients from each cohort will be combined for the summaries. If there is a clear increase in AE rates for placebo patients across the cohorts, the AEs will also be summarized by cohort.

AEs will be summarized by counts and percentages of patients by treatment group. Laboratory data and vital signs will be summarized by treatment group as summary statistics for value and change from baseline at each individual time point. Summary statistics will include n, arithmetic mean, median, arithmetic SD, minimum, and maximum.

Additional safety parameters will be analyzed descriptively by treatment group. Descriptive statistics (n, mean, standard deviation (SD), median, minimum, maximum) will be calculated by treatment group and time point for continuous variables. Frequencies and percentages will be presented by treatment group for categorical and ordinal variables.

### 9.2.5.2 Data Monitoring Committee

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for anti-IL-21 mAb. The recommendations made by the DMC (ie, dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will

forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.

The DMC will have access to unblinded treatment information during the clinical trial. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of an anti-IL-21 mAb treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.

### 9.2.6 Pharmacokinetic and Pharmacodynamic Data

# 9.2.6.1 Analysis of Pharmacokinetic Data

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:

- A listing of all plasma BOS161721 concentrations by patient at actual times post dose;
- A descriptive summary of plasma BOS161721 concentrations. Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.

Details will be available in the SAP.

#### 9.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Binary PD endpoints will be assessed for the FAS population. Binary PD endpoints will be assessed via CMH analysis. Continuous PD endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-by-time interaction, baseline covariate, and covariate-by-time interaction. Normality will be assessed via diagnostic residual plots and Shapiro-Wilk statistic, but not as a formal statistical test of normality. If substantial departures from normality are observed, transformation will be used (eg, log and/or rank).

Details will be available in the SAP.

### 9.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints.

Details will be available in the SAP.

# 9.3 Interim Analysis and Power

Two IAs are planned for this study. The initial IA will be conducted at the time of the POC decision for dose selection.

The second IA will be performed for futility. IA2 is planned to be conducted at Day 90 when SRI-4 response is determined for approximately 60 patients (including all patients at the same dose level/matching placebo from the MAD study) after completing 3 months of treatment. The purpose of the IA2 is to assess if the trial could stop for an early futility conclusion, or continue. Since there is no plan to stop the trial for an early efficacy conclusion, there is no impact on the type 1 error. If that intention changes, then p < 0.0001 is required for an early efficacy conclusion at the IA2 in order to not impact the planned type 1 error level.

Nominal time profiles will be used for calculating PK parameters in the IA2. Details will be available in the SAP.

### 10 ETHICS AND RESPONSIBILITIES

#### 10.1 Good Clinical Practice

The procedures set out in this protocol are designed to ensure that the sponsor and the principal investigator abide by the principles of the International Council for Harmonisation (ICH) guidelines on GCP and the Declaration of Helsinki (Version 2013). The clinical study also will be carried out in the keeping with national and local legal requirements (in accordance with US IND regulations [21 CFR 56]).

#### 10.2 DMC

The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) suggest dose for POC portion of the study.

The DMC considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

# 10.3 Institutional Review Board/Independent Ethics Committee

Independent Ethics Committees (IEC)/Institutional Review Boards (IRB) must meet the guidelines set out by the U.S. Food and Drug Administration (FDA) and conform to local laws and customs where appropriate. Written IRB/IEC approval for the protocol and the signed ICF must be obtained and transmitted to Boston Pharmaceuticals or representative before the study can be initiated. The IRB/IEC must be informed of and approve all protocol amendments. The investigator will ensure that this study is conducted in full conformance with all applicable local and regional laws and regulations. The complete text of the World Medical Association Declaration of Helsinki is given in APPENDIX 2.

#### **10.4** Informed Consent

Before each patient undergoes any protocol required assessments or procedure, the written informed consent will be obtained according to the regulatory and legal requirements of the participating country. As part of this procedure, the principal investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study patient should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The principal investigator or designee will provide the sponsor with a copy of the IRB-approved ICF prior to the start of the study.

The informed consent document must be signed and dated; 1 copy will be handed to the patient and the principal investigator will retain a copy as part of the clinical study records. The principal investigator will not undertake any investigation specifically required for the clinical study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented.

If the informed consent document is revised, it must be reviewed and approved by the responsible IRB/IEC. Patients currently enrolled may need to sign this revision (based on IRB/IEC requirements) and all future subjects enrolled in the clinical study will be required to sign this revised ICF.

# 10.5 Records Management

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes. The principal investigator or designee will cooperate with the sponsor's representative(s) for the periodic review of study documents to ensure the accuracy and completeness of the data capture system at each scheduled monitoring visit.

Electronic consistency checks and manual review will be used to identify any errors or inconsistencies in the data. This information will be provided to the respective study sites by means of electronic or manual queries.

The principal investigator or designee will prepare and maintain adequate and accurate study documents (medical records, ECGs, AE and concomitant medication reporting, raw data collection forms, etc.) designed to record all observations and other pertinent data for each patient receiving BOS161721 or placebo.

The principal investigator will allow sponsor representatives, contract designees, authorized regulatory authority inspectors, and the IRB to have direct access to all documents pertaining to the study.

Electronic case report forms are required and should be completed for each randomized patient. It is the principal investigator's responsibility to ensure the accuracy, completeness, legibility, and timeliness of the data reported on the patients' eCRF. Electronic case report forms should be completed in a timely fashion to support the study timelines. Source documentation supporting the eCRF data should indicate the patient's participation in the study and should document the dates and details of study procedures, AEs, and patient status. The principal investigator or designated representative should complete and the principal investigator should verify the source documents as the information is collected. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the Sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes.

#### **10.6** Source Documentation

The documents that will form the source data for the clinical study (eg, patient charts, laboratory reports) must be defined and documented in the in-house study master file prior to the start of the study. Data on the eCRFs which will be checked against source data during monitoring visits must also be defined and documented in the in-house study master file including the percentage of each of the source data to be verified and the percentage of patients' eCRFs to be monitored.

# 10.7 Study Files and Record Retention

According to ICH guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of BOS161721. However, these documents should be retained for a longer period if required by the applicable legal requirements.

### 11 AUDITING AND MONITORING

Throughout the course of the study, the study monitor will make frequent contacts with the investigator. This will include telephone calls and on-site visits. The study will be routinely monitored to ensure compliance with the study protocol and the overall quality of data collected. During the on-site visits, the eCRFs will be reviewed for completeness and adherence to the protocol. As part of the data audit, source documents will be made available for review by the
study monitor. The study monitor may periodically request review of the investigator study file to assure the completeness of documentation in all respects of clinical study conduct. The study monitor will verify that each patient has proper consent documentation from the patient and/or patient's authorized representative for study procedures and for the release of medical records to the sponsor, FDA, other regulatory authorities, and the IRB. The study monitor will also verify that assent was obtained for patients not capable of providing informed consent or that documentation is provided by the investigator explaining why the patient was unable to provide assent. The investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the investigator will permit inspection of the study files by authorized representatives of the regulatory agencies. On completion of the study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

Throughout the course of the study, the medical monitor will determine eligibility of all screened patients, will address any medical issues that might arise, clarify medical questions, review patient safety data (eg, AE/SAE, laboratory, and ECG), and partner with the study team in the overall study management. The study medical monitoring plan will document additional details of the study medical oversight and monitoring.

#### 12 AMENDMENTS

Protocol modifications, except those intended to reduce immediate risk to study patients, may be made only by Boston Pharmaceuticals. A protocol change intended to eliminate an apparent immediate hazard to patients may be implemented immediately, provided the IRB/IEC is notified within 5 days.

Any permanent change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB/IEC and the investigator must await approval before implementing the changes. Boston Pharmaceuticals will submit protocol amendments to the appropriate regulatory authorities for approval.

If in the judgment of the IRB/IEC, the investigator, and/or Boston Pharmaceuticals, the amendment to the protocol substantially changes the study design and/or increases the potential risk to the patient and/or has an impact on the patient's involvement as a study participant, the currently approved written ICF will require similar modification. In such cases, informed consent will be renewed for patients enrolled in the study before continued participation.

#### 13 STUDY REPORT AND PUBLICATIONS

Boston Pharmaceuticals is responsible for preparing and providing the appropriate regulatory authorities with clinical study reports according to the applicable regulatory requirements.

By signing the protocol, the principal investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the principal investigator's name, address, qualifications, and extent of involvement.

The principal investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted and obtained approval from the sponsor in advance.

#### 14 STUDY DISCONTINUATION

Both Boston Pharmaceuticals and the principal investigator reserve the right to terminate the study at the investigator's site at any time. Should this be necessary, Boston Pharmaceuticals or a specified designee will inform the appropriate regulatory authorities of the termination of the study and the reasons for its termination, and the principal investigator will inform the IRB/IEC of the same. In terminating the study Boston Pharmaceuticals and the principal investigator will assure that adequate consideration is given to the protection of the patients' interests.

#### 15 CONFIDENTIALITY

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from Boston Pharmaceuticals, except to the extent necessary to obtain informed consent from patients who wish to participate in the trial or to comply with regulatory requirements. However, authorized regulatory officials, IRB/IEC personnel, Boston Pharmaceuticals, and its authorized representatives are allowed full access to the records.

Identification of patients and eCRFs shall be by initials, birthdate, or patient number. Documents that identify the patient (eg, the signed informed consent document) must be maintained in confidence by the principal investigator. If required, the patient's full name may be made known to an authorized regulatory agency or other authorized official.

#### 16 REFERENCES

1 Urowitz MB, Gladman DD. How to improve morbidity and mortality in systemic lupus erythematosus. Rheumatology 2000;39:238-44.

- 2 Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, et al. Morbidity and Mortality in Systemic Lupus Erythematosus During a 10-Year Period. Medicine 2003;82(5):299-308.
- 3 Pons-Estel GJ, Alarcón GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010;39(4):257. Epub 2009 Jan 10.
- 4 Kanta H, Mohan C. Three Checkpoints in lupus development: central tolerance in adaptive immunity, peripheral amplification by innate immunity, and end-organ inflammation. Genes and Immunity 2009;10:390-6.
- 5 Dall'Aqua WF, Kiener PA, Wu H. Properties of Human IgG1s Engineered for Enhanced Binding to the Neonatal Fc Receptor (FcRn). J Biol Chem. 2006 Aug 18, 281(33):23514-24.
- 6 Spolski R, Leonard WJ. The Yin and Yang of interleukin-21 in allergy, autoimmunity and cancer. Curr Opin Immunol. 2008a;20:295-301.
- 7 Asao H, Okuyama C, Kumaki S, Ishii N, Tsuchiya S, Foster D, et al. Cutting edge: the common gamma-chain is an indispensable subunit of the IL-21 receptor complex. J Immunol. 2001;167:1-5.
- 8 Habib T, Senadheera S, Weinberg K, Kaushansky K. The common gamma chain (gamma c) is a required signaling component of the IL-21 receptor and supports IL-21-induced cell proliferation via JAK3. Biochemistry. 2002;41:8725-31.
- 9 Spolski R, Leonard WJ. Interleukin-21: basic biology and implications for cancer and autoimmunity. Annu Rev Immunol. 2008b;26:57-79.
- 10 Puga I, Cols M, Barra CM, He B, Cassis L, Gentile M, et al. B-cell-helper neutrophils stimulate the diversification and production of immunoglobulin in the marginal zone of the spleen. Nat Immunol. 2011;13(2):170-80.
- 11 Costanzo A, Chimenti MS, Botti E, Caruso R, Sarra M, Monteleone G. IL-21 in the pathogenesis and treatment of skin diseases. J Dermatol Sci. 2010;60(2):61-6.
- 12 Avery DT, Bryant VL, Ma CS, de Waal Malefy R, Tangye SG. IL-21-induced isotype switching to IgG and IgA by human naive B cells is differentially regulated by IL-4. J Immunol. 2008;181:1767-79.
- 13 Rasmussen TK, Andersen T, Bak, RO, Yiu G, Sorensen CM, Stengaard-Pedersen K, et al. Overexpression of microRNA-155 increases IL-21 mediated STAT3 signaling and IL-21 production in systemic lupus erythematosus. Arthritis Research & Therapy 2015;17(154)

and disease. Immunol Rev. 2008;223:60-86.

- 14 Ettinger R, Kuchen S, Lipsky PE. The role of IL-21 in regulating B-cell function in health
- 15 Caprioli F, Sarra M, Caruso R, Stolfi C, Fina D, Sica G, et al. Autocrine regulation of IL-21 production in human T lymphocytes. J Immunol. 2008;180(3):1800-7.
- 16 Yang L, Anderson DE, Baecher-Allan C, Hastings WD, Bettelli E, Oukka M, et al. IL-21 and TGF-beta are required for differentiation of human T(H)17 cells. Nature. 2008;454(7202):350-2.
- 17 Tangye SG, Ma CS, Brink R, Deenick EK. The good, the bad and the ugly TFH cells in human health and disease. Nat Rev Immunol. 2013;13(6):412-26.
- 18 Fantini MC, Rizzo A, Fina D, Caruso R, Becker C, Neurath MF, et al. IL-21 regulates experimental colitis by modulating the balance between Treg and Th17 cells. Eur J Immunol. 2007;37(11):3155-63.
- 19 Peluso I, Fantini MC, Fina D, Caruso R, Boirivant M, MacDonald TT, et al. IL-21 counteracts the regulatory T-cell-mediated suppression of human CD4+ T lymphocytes. J Immunol. 2007;178(2):732-9.
- 20 Hippen KL, Bucher C, Schirm DK, Bearl AM, Brender T, Mink KA, et al. Blocking IL-21 signaling ameliorates xenogeneic GVHD induced by human lymphocytes. Blood. 2012;119(2):619-28.
- 21 Davis ID, Skrumsager BK, Cebon J, Nicholaou T, Barlow JW, Moller NP, et al. An open-label, two-arm, phase I trial of recombinant human interleukin-21 in patients with metastatic melanoma. Clin Cancer Res. 2007;13:3630-6.
- 22 Frederiksen KS, Lundsgaard D, Freeman JA, Hughes SD, Holm TL, Skrumsager BK, et al. IL-21 induces in vivo immune activation of NK cells and CD8(+) T-cells in patients with metastatic melanoma and renal cell carcinoma. Cancer Immunol Immunother. 2008;57(10):1439-49.
- 23 Karrich JJ, Jachimowski LC, Nagasawa M, Kamp A, Balzarolo M, Wolkers MC, et al. IL-21- stimulated human plasmacytoid dendritic cells secrete granzyme B, which impairs their capacity to induce T-cell proliferation. Blood. 2013;121(16):3103-11.
- 24 Lindner S, Dahlke K, Sontheimer K, Hagn M, Kaltenmeier C, Barth TF, et al. Interleukin-21-induced granzyme B-expressing B-cells infiltrate tumors and regulate T-cells. Cancer Res. 2013;73(8):2468-79.
- 25 Monteleone G, Caruso R, Fina D, Peluso I, Gioia V, Stolfi C, et al. Control of matrix metalloproteinase production in human intestinal fibroblasts by interleukin 21. Gut. 2006;55(12):1774-80.
- 26 Nakou M, Papadimitraki ED, Fanouriakis A, Bertsias GK, Choulaki C, Goulidaki N, et al. Interleukin-21 is increased in active systemic lupus erythematosus patients and contributes to the generation of plasma B-cells. Clin Exp Rheumatol. 2013;31(2):172-9.

- 27 Li Q, Liu Z, Dang E, Jin L, He Z, Yang L, et al. Follicular helper T-cells (Tfh) and IL-21 involvement in the pathogenesis of bullous pemphigoid. PLoS One. 2013;8(7):e68145.
- 28 Liu R, Wu Q, Su D, Che N, Chen H, Geng L, et al. A regulatory effect of IL-21 on T follicular helper-like cell and B-cell in rheumatoid arthritis. Arthritis Res Ther. 2012;14(6):R255.
- 29 Kang KY, Kim HO, Kwok SK, Ju JH, Park KS, Sun DI, et al. Impact of interleukin-21 in the pathogenesis of primary Sjögren's syndrome: increased serum levels of interleukin-21 and its expression in the labial salivary glands. Arthritis Res Ther. 2011;13(5):R179.
- 30 Terrier B, Geri G, Chaara W, Allenbach Y, Rosenzwajg M, Costedoat-Chalumeau N, et al. Interleukin-21 modulates Th1 and Th17 responses in gianT-cell arteritis. Arthritis Rheum. 2012a;64(6):2001-11.
- 31 Terrier B, Costedoat-Chalumeau N, Garrido M, Geri G, Rosenzwajg M, Musset L, et al. Interleukin 21 correlates with T-cell and B-cell subset alterations in systemic lupus erythematosus. J Rheumatol. 2012b;39(9):1819-28.
- 32 International Conference on Harmonisation. Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals S6 (R1). 2011.
- 33 Wang W, Wang EQ, Balthasar JP. Monoclonal Antibody Pharmacokinetics and Pharmacodynamics. Clin Pharm & Ther 2008; 84(5):548-58.
- 34 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 35 Elsaesser H, Sauer K, Brooks DG. IL-21 is required to control chronic viral infection. Science. 2009;324(5934):1569-72
- 36 Kotlarz D, Zietara N, Uzel G, Weidemann T, Braun CJ, Diestelhorst J, et al. Loss-of-function mutations in the IL-21 receptor gene cause a primary immunodeficiency syndrome. J Exp Med. 2013;210(3):433-43.
- 37 Hunter PR, Nichols G. Epidemiology and clinical features of Cryptosporidium infection in immunocompromised patients. Clinical microbiology reviews. 2002;15(1):145-54.
- 38 Desjardins M, Mazer BD. B-cell memory and primary immune deficiencies: interleukin-21 related defects. Curr Opin Allergy Clin Immunol. 2013;13(6):639-45.
- 39 Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. *Nephron*. 1976;16(1):31-41.
- 40 Guidelines for Using the QuantiFERON®-TB Gold Test for Detecting Mycobacterium tuberculosis Infection, US: http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5415a4.htm.

- 41 NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, available at https://evs.nci.nih.gov/ftp1/CTCAE/About.html.
- 42 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 43 Posner K, Melvin G a, Stanley B, Oquendo M a, Gould M. Factors in the assessment of suicidality in youth. *CNS Spectr*. 2007;12(2):156-162.
- 44 Castrejon I, Tani C, Jolly M, Huang A, Mosca M. Indices to assess patients with systemic lupus erythematosus in clinical trials, long-term observational studies, and clinical care. Clin Exp Rheumatol 2014; 32(85):S85-95.
- 45 Furie R, Wang L, Drappa J, Illei G. Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] Response Is Associated with Global Benefit in Patients with Moderate to Severe SLE [abstract]. *Arthritis Rheumatol.* 2016; 68 (suppl 10).
- 46 Thanou A, Chakravarty E, James JA, Merrill JT. Which outcome measures in SLE clinical trials best reflect medical judgment? Lupus Science & Medicine 2014;1:e000005. doi:10.1136/lupus-2013-000005.
- 47 Wallace DJ, Kalunian K, Petri MA, Strand V, Houssiau FA, Pike M, et al. Efficacy and safety of epratuzumab in patients with moderate/severe active systemic lupus erythematosus: results from EMBLEM, a phase IIb, randomised, double-blind, placebo-controlled, multicentre study. *Ann Rheum Dis* 2014;73:183-90.
- 48 Albrecht J, Taylor L, Berlin JA, Dulay S, Ang G, Fakharzadeh S. The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index): An Outcome Instrument for Cutaneous Lupus Erythematosus. J Invest Derm. 2005;125(5):889-94.
- 49 Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is Valid, and Renal and Pulmonary Organ Scores are Predictors of Sever Outcome in Patients with Systemic Lupus Erythematosus. Br J Rheumatol. 1996;35:248-54.



#### 17 APPENDICES

#### APPENDIX 1 NAMES OF STUDY PERSONNEL

Sponsor: Boston Pharmaceuticals

55 Cambridge Parkway Suite 401 Cambridge, MA 02142, USA

Medical Monitor:

PPD

PPD

Clinical Research Organizations:

PPD

PPD

Bioanalytical Laboratory:

PPD

**PPD** 

Central Laboratory:

#### APPENDIX 2 DECLARATION OF HELSINKI

#### WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI

Ethical Principles
For
Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly
Helsinki, Finland, June 1964
and amended by the
29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
and the

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### A. INTRODUCTION

The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.

It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.

The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my subject will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the subject's interest when providing medical care which might have the effect of weakening the physical and mental condition of the subject."

Medical progress is based on research, which ultimately must rest in part on experimentation involving human subjects.

In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.

The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic, and therapeutic procedures and the understanding of the etiology and pathogenesis of disease. Even the best-proven prophylactic, diagnostic, and therapeutic methods must continuously be challenged through research for their effectiveness, efficiency, accessibility, and quality.

In current medical practice and in medical research, most prophylactic, diagnostic, and therapeutic procedures involve risks and burdens.

Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.

Research investigators should be aware of the ethical, legal, and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal, or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### B. BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.

Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.

Appropriate caution must be exercised in the conduct of research, which may affect the environment, and the welfare of animals used for research must be respected.

The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any SAEs. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.

The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles enunciated in this Declaration.

Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a subject of the research, even though the subject has given consent.

Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the

subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.

Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.

Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.

Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.

The subjects must be volunteers and informed participants in the research project.

The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the subject's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.

In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.

When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.

For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the investigator must obtain informed consent from the legally authorized representative in accordance with applicable law. These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.

When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the investigator must obtain that assent in addition to the consent of the legally authorized representative.

Research on individuals from whom it is not possible to obtain consent, including proxy or advance consent, should be done only if the physical/mental condition that prevents obtaining

informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.

Both authors and publishers have ethical obligations. In publication of the results of research, the investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic, or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the subjects who are research subjects.

The benefits, risks, burdens, and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic, or therapeutic method exists.

At the conclusion of the study, every subject entered into the study should be assured of access to the best-proven prophylactic, diagnostic, and therapeutic methods identified by the study.

The physician should fully inform the subject which aspects of the care are related to the research. The refusal of a subject to participate in a study must never interfere with the subject-physician relationship.

In the treatment of a subject, where proven prophylactic, diagnostic, and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the subject, must be free to use unproven or new prophylactic, diagnostic, and therapeutic measures, if in the physician's judgment it offers hope of saving life, re-establishing health, or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases, new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.

# APPENDIX 3 COMMONLY USED CORTICOSTEROID EQUIVALENTS

| Medication | Dose Equivalence |
|--------------------|------------------|
| Prednisone | 20 mg |
| Cortisone | 100 mg |
| Hydrocortisone | 80 mg |
| Prednisolone | 20 mg |
| Methylprednisolone | 16 mg |
| Triamcinolone | 16 mg |
| Budesonide | 4 mg |
| Dexamethasone | 3 mg |
| Bethamethasone | 2.4 mg |

#### APPENDIX 4 MEDICATION WASHOUT PERIODS

#### WASHOUT TIMES OF MEDICATIONS BASED ON 5 HALF-LIVES

| Medication | Discontinuing Prior to Signing Consent |
|---|---|
| Abatacept (CTLA4Ig) | 24 weeks |
| Alefacept | 12 weeks |
| AMG 623 (blisibimod) | 24 weeks |
| Anifrolumab | 12 weeks |
| Atacicept (TACI-Ig) | 12 weeks |
| Belimumab | 48 weeks |
| Cyclophosphamide | 24 weeks |
| Cyclosporine (except for CSA eye drops) | 4 weeks |
| Danazol | 4 weeks |
| Dapsone | 4 weeks |
| Eculizumab | 12 weeks |
| Efalizumab | 12 weeks |
| Epratuzumab | 24 weeks |
| Intravenous globulin | 4 weeks |
| Leflunomide | 8 weeks (4 weeks for washout with cholestyramine) |
| Lenalidomide with cholestiramine | 8 weeks |
| Lupuzor | 12 weeks |
| Memantine | 4 weeks |
| Natalizumab | 24 weeks |
| Ocrelizumab | 48 weeks (or 24 weeks with recovery of B cell) |
| Pimecrolimus | 4 weeks |
| Plasmapheresis | 24 weeks |
| Retinoids (oral or topical) | 4 weeks |
| Rituximab | 48 weeks (or 24 weeks with recovery of B cell) |
| Sirolimus | 4 weeks |
| Tacrolimus | 4 weeks |
| Thalidomide | 8 weeks |
| Tocilizumab | 12 weeks |

## APPENDIX 5 BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA)





# A RANDOMIZED DOUBLE-BLIND PHASE 1b/2 COMBINED STAGGERED MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF LIMITED STANDARD OF CARE

**SPONSOR** Boston Pharmaceuticals, Inc.

55 Cambridge Parkway, Suite 401

Cambridge, MA 02142

United States of America (USA)

INVESTIGATIONAL COMPOUND: BOS161721

PROTOCOL NUMBER: BOS161721-02

PHASE Phase 1b/2

INVESTIGATIONAL NEW DRUG (IND)

**NUMBER:** 

131796


**VERSION NUMBER:** V1.0

**VERSION DATE:** 06 October 2017

BOS161721 Boston Pharmaceuticals, Inc.

Clinical Study Protocol: BOS161721-02

#### CLINICAL PROTOCOL APPROVAL FORM

Protocol Title: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

Study No: BOS161721-02

Original Protocol Date: 05 October 2017

Protocol Version No: v1.0

Protocol Version Date: 06 October 2017

This study protocol was subject to critical review and has been approved by sponsor. The information contained in this protocol is consistent with:

- The current risk-benefit evaluation of the investigational product.
- The moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (APPENDIX 2), and principles of Good Clinical Practices (GCP) as described in 21 Code of Federal Regulations (CFR) parts 50, 54, 56 and 312 and according to applicable local requirements.

The investigator will be supplied with details of any significant or new findings, including adverse events, relating to treatment with the investigational product.

I agree with these statements and indicate my approval by signature for this protocol:

| Name and Title | Signature | Date |
|---|---|---|
| PPD , MD Vice President, Clinical Development Boston Pharmaceuticals | PPD | 10/6/2017 |
| PPD Clinical Operations Lead Boston Pharmaceuticals | PPD | 10/6/2017 |
| PPD , MD, PhD Vice President, Clinical Development and Safety Officer Boston Pharmaceuticals | PPD | 10/6/2017 |

#### BOS161721-02

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

#### CONFIDENTIALITY AND INVESTIGATOR STATEMENT

The information contained in this protocol and all other information relevant to BOS161721 are the confidential and proprietary information of Boston Pharmaceuticals, Inc., and except as may be required by federal, state, or local laws or regulation, may not be disclosed to others without prior written permission of Boston Pharmaceuticals, Inc.

I have read the protocol, including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described. I will conduct this study as outlined herein, in accordance with the regulations stated in the Federal Code of Regulations for Good Clinical Practices and International Council for Harmonisation (ICH) guidelines, and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and any amendments, and access to all information provided by Boston Pharmaceuticals, Inc., or specified designees. I will discuss the material with them to ensure that they are fully informed about BOS161721 and the study.

| Principal Investigator Name (printed) | | Signature |
|---------------------------------------|-----------------|-----------|
| | — — Site Number | |


#### PROTOCOL SUMMARY

Title:

A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care

Indication

Adults with moderately to severely active SLE

Background and Rationale

SLE is a chronic systemic autoimmune disease with considerable heterogeneity in clinical manifestations and disease course. There is evidence that B- and T-cells are critical to the development of the disease, and that T-cell-derived cytokines such as interleukin-21 (IL-21) are involved in the SLE-associated inflammatory pathological response.

BOS161721 is a humanized immunoglobulin G1 (IgG1) triple mutation monoclonal antibody (mAb) intended to have an extended terminal elimination half-life ( $t_{1/2}$ ) that selectively binds to and neutralizes IL-21, which acts on multiple cell types that drive inflammation and autoimmunity. In vivo, BOS161721 inhibits T-cell dependent antigen responses of B-cells and is being developed as a potential treatment for adults with moderately to severely active SLE.

Nonclinical studies have evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), pharmacokinetics (PK), and immunogenicity of BOS161721 administered intravenously (IV) and subcutaneously (SC). The no observed adverse effect levels (NOAELs) in Cynomolgus monkeys were determined to be 100 mg/kg IV and 50 mg/kg SC, the highest doses tested. No SC animals had injection reactions.

In a Phase 1 single ascending dose (SAD) study, BOS161721 was administered IV and SC to healthy male and female adult subjects. This double-blind, placebo-controlled study evaluated 8 ascending dose levels (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) for safety, tolerability, PK, PD and immunogenicity. Overall, there were no clinically significant safety or tolerability findings from this study.

Results from the Phase 1 SAD study informed the dose regimens used for the multiple ascending doses (MAD) Phase 1b study in this trial. The MAD study will involve 3 cohorts. The Phase 2 portion will be a proof of concept (POC) study, where dose selection will be based on the sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD study of


30 patients treated with BOS161721/placebo. The purpose of the study is to establish safe and effective dosages for adult patients with moderately to severely active SLE.

#### **Objectives:**

#### **MAD Phase 1b Study**

#### **Primary Objective:**

To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20 mg, 60 mg, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose.

#### **POC Phase 2 Study**

#### **Primary Objective:**

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on the SLE Responder Index 4 (SRI-4), with sustained reduction of oral corticosteroids (CS), in adult patients with moderately to severely active SLE on limited background standard of care treatment.

#### **Secondary Objectives:**

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment, including:

- Changes in SLE-specific autoantibody titers;
- Changes in complement 3 and 4 (C3 and C4) levels;
- Responses on SRI-4, SLE Responder Index 5 and 6 (SRI-5, and SRI-6), with sustained reduction of oral CS;
- Response on the British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (BICLA);
- Response on the Cutaneous Lupus Erythematosus Area and Severity Index (CLASI);
- Changes in the SLE Disease Activity Index 2000 (SLEDAI-2K);
- Changes in the American College of Rheumatology (ACR)-28 joint count.

Confidential

BOS161721 Boston Pharmaceuticals, Inc. Clinical Study Protocol: BOS161721-02

#### **Endpoints:**

#### **Phase 1b MAD Study**

#### **Primary Endpoints:**

Evaluation of safety, tolerability, and immunogenicity at each dose level, to determine the optimal dose, will include the recording of the following parameters:

- Incidence and severity of adverse events (AEs) and serious adverse events (SAEs);
- 12-lead electrocardiograms (ECGs);
- Vital signs (blood pressure [BP], heart rate, and temperature);
- Clinical laboratory assessments;
- Physical examinations;
- Evaluation for anti-drug antibodies (ADAs).

#### **Exploratory Endpoints:**




#### **Other Endpoints:**



#### **PRO Endpoints:**



#### **Phase 2 POC Study**

#### **Primary Efficacy Endpoint:**

The primary efficacy endpoint is the proportion of patients who achieve treatment response as measured by the SRI-4 at Week 28, along with a sustained reduction of oral CS ( $\leq$  10 mg/day and  $\leq$  Day 1 dose) between Week 16 and Week 28.

#### **Secondary Efficacy Endpoints:**

- The proportion of patients who achieve treatment response for the SRI-5 and SRI-6 at Week 28, along with a sustained reduction of oral CS (≤ 10 mg/day and ≤ Day 1 dose) between Week 16 and Week 28;
- Changes from baseline in dsDNA, ANA, SSA, SSB, RNP, Sm, APL autoantibodies, at Week 16 and Week 28;
- Changes from baseline in C3 and C4 levels at Week 16 and Week 28;
- Changes from baseline in the SLEDAI-2K at Week 28;
- Time to BILAG A or B flare;
- Changes from baseline in the CLASI at Week 28;
- The proportion of patients with a BICLA response at Week 28;

- The proportion of patients with CLASI response at Week 28;
- Changes from baseline (percentage) in swollen joints and tender joints ACR-28 joint count;
- Assessment of safety, tolerability, and immunogenicity as described for the primary endpoint in the MAD Phase 1b study.

#### **Exploratory Endpoints:**



#### **Other Endpoints:**

- CCI
- CCI
- CCI

#### **PRO Endpoints:**

- CCI
- CCI

#### **Study Design:**

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of multiple SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly. The trial will consist of a staggered MAD Phase 1b and POC Phase 2 studies. Both studies will be double-blinded with each patient having the same number of doses (7), and visits; the duration will be 180 days, followed by a 90-day follow-up safety observation period.

The MAD Phase 1b study phase will consist of 3 cohorts, with Cohort 1 containing 6 patients, where 5 of these patients will receive

BOS161721 (active), and 1 will receive placebo. Cohorts 2 and 3 will each contain 12 patients, including 9 active and 3 placebo patients. Dose selection for each cohort is based on 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. Each of the 3 doses (20 mg, 60 mg, and 120 mg) selected for the MAD study are projected not to exceed the mean peak levels or exposures of that achieved in the SAD study following the single 240 mg SC dose. Each patient may receive a total of 7 SC monthly doses on Days 1, 30, 60, 90, 120, 150, and 180.

The MAD study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after a data monitoring committee [DMC] evaluates the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing (based on the dose level determined after DMC evaluation of the safety and tolerability data from Cohort 2 and Cohort 1). Two weeks after the last patient in Cohort 3 receives the second dose, the DMC will conduct a data review for the first interim analysis (IA1) to determine which dose will be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available when the last patient in Cohort 3 reaches 60 days (dose 2). Once the POC dose decision has been made, screening for the POC study can begin.

For the POC study, 156 patients will be randomized to active or placebo groups in a 2:1 ratio. As in the MAD study, each patient in the POC study may receive a total of 7 SC monthly doses on Days 1, 30, 60, 90, 120, 150, and 180. A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 1 (randomization day). One oral CS "burst" for increased SLE disease activity may occur during the study either between Weeks 1 and 8 or between Weeks 16 and 20. Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits. Tapering may occur after randomization except within 8 weeks of the primary (Week 28) and secondary (Week 16) endpoint assessments. Between Week 8 and Week 16, and between Week 20 and Week 28, oral corticosteroid (OCS) doses must be held constant otherwise the patient will be declared a

non-responder in efficacy assessments.

Data from 60 patients, including the 12 from the MAD study, or 6 fewer if the low dose is chosen, who are in the cohort of the chosen dose for the POC study who complete 3 months of treatment will be used in a second IA (IA2) at Week 16 to assess if the trial could stop for an early futility conclusion. If futility is not claimed in the IA2, the POC study will continue to 156 patients.

Following the 6-month treatment period, primary and secondary efficacy endpoints will be assessed for each patient, after providing their 24-week disease activity assessments. DMC monitoring will be conducted periodically throughout the study as described in the DMC charter.

# Main Criteria for Inclusion and Exclusion

#### **Inclusion Criteria:**

- 1. Men and women, ages 18 to 70 years, inclusive.
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion OR Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously.
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated ANA  $\geq$  1:80 via immunofluorescent assay at the central laboratory;
  - b. Positive anti-dsDNA or anti-Sm above the normal level as determined by the central laboratory;
  - c. C3 or C4 below normal as determined by the central lab.
- 5. At screening, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory

- results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia);
- ii. Points from lupus headache and organic brain syndrome will also be excluded.
- 6. On Day 1, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis.
    - i. Excluding parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia and leukopenia;
    - ii. Points from lupus headache and organic brain syndrome are also excluded.
- 7. Patients must have at least 1 of the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system;
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis as defined in the protocol Section 5.4;
  - c. If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores.
- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX).
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must

be stable at a maximum of 10 mg/day for at least 5 days prior to Day 1 (randomization).

- 9. Women of childbearing potential (WOCBP; see Section 5.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose.
  - b. Must not be breastfeeding;
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS1617219 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion;
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion.
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures.

#### **Exclusion Criteria**

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE;
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE);
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed.
- 3. Any major surgery within 6 weeks of study drug administration, (Day 1), or any elective surgery planned during the course of the study:
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB;

- b. History of active TB;
- c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 1 and continues to receive the prophylactic treatment during study until the treatment course is completed.
- Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed;
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS;
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary
  - a. However, treatment for asthma with inhalational CS therapy is allowed.
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study;
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic antibiotics or hospitalization;
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years;
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness;
- 12. Cryptosporidium in the stool sample at screening;
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening;
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening;

- 15. CD4+ count  $< 500/\mu$ L at screening;
- 16. Platelets  $< 50,000/\text{mm}^3$  (50  $\times$  10<sup>9</sup>/L) or  $< 35,000/\text{ mm}^3$  (35  $\times$  10<sup>9</sup>/L) if related to SLE, at screening;
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if due to anemia related to SLE.
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol);
- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation;
- 20. Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) > 2 × the upper limit of normal (ULN) at screening, unless explicitly related to lupus based on the investigator's judgment;
- 21. Creatinine kinase (CK) > 3.0  $\times$  ULN at screening unless related to lupus myositis.
- 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome);
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study;
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic mAb (eg, IgG protein) or molecules made of components of mAbs;
- 25. History substance and/or alcohol abuse, or dependence within the past 1 year, at the investigator's judgement;
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision;
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are

- employees of the sponsor or directly involved in the conduct of the trial;
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer;
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 on the Columbia Suicide severity Rating Scale (C-SSRS);
- 31. Current or pending incarceration;
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Below is a summary of the statistical methods. Further details can be found in Section 9.

Baseline and patient characteristics will be summarized via appropriate summary statistics by treatment group and overall, for each phase of the trial.

Binary efficacy endpoints will be compared between treatments via Cochran-Mantel-Haenszel (CMH) analysis. Continuous efficacy endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-by-time interaction, baseline covariate, and covariate-by-time interaction. Summary statistics will be provided by dose/treatment for all safety endpoints. Details will be provided in the statistical analysis plan (SAP).

Two IAs are planned for this study. The initial IA (IA1) will be conducted at the time of the POC decision for dose selection. The second IA (IA2) will be performed for futility. IA2 is planned to be conducted when SRI-4 response is determined for approximately 60 patients (including all patients at the same dose level/matching placebo from the MAD study) after completing 3 months of treatment. The purpose of IA2 is to assess if the trial could stop for an early futility conclusion, or continue. Since there is no plan to stop the trial for an early efficacy conclusion, there is no impact on the type 1 error level.

AEs will be summarized by counts and percentages of patients by treatment group. Laboratory data and vital signs will be summarized by treatment group as summary statistics for value and change from baseline at each individual time point. Summary statistics will include n, arithmetic mean, median, arithmetic SD, minimum, and maximum.

#### Statistical Considerations

The PK parameter data will be listed and summarized descriptively in tabular format. Binary PD endpoints will be assessed for the full analysis set (FAS) population via CMH analysis. Continuous PD endpoints will be assessed via ANCOVA repeated measures mixed model analysis with multiple factors. PK and PD relationships will be explored graphically and where appropriate model based methods of analysis will used.

## TABLE OF CONTENTS

| A RANDOMIZED DOUBLE-BLIND PHASE 1B/2 COMBINED STAGGERED | |
|---------------------------------------------------------|----|
| MULTIPLE DOSE ESCALATION STUDY OF BOS161721 IN SYSTEMIC | |
| LUPUS ERYTHEMATOSUS (SLE) PATIENTS ON A BACKGROUND OF | |
| LIMITED STANDARD OF CARE | |
| CLINICAL PROTOCOL APPROVAL FORM | |
| CONFIDENTIALITY AND INVESTIGATOR STATEMENT | |
| PROTOCOL SUMMARY | |
| TABLE OF CONTENTS | |
| LIST OF IN-TEXT TABLES | |
| LIST OF IN-TEXT FIGURES | |
| LIST OF ABBREVIATIONS | |
| 1 INTRODUCTION AND RATIONALE | |
| 1.1 Indication | |
| 1.2 Background and Rationale | |
| 1.2.1 Overview of the Disease State | 27 |
| 1.2.2 BOS161721 Development | 27 |
| 1.2.2.1 Interleukin-21 | 28 |
| 1.2.2.2 Preclinical Studies | 29 |
| 1.2.2.3 Clinical Studies | |
| 1.2.3 Study Dose Selection | 31 |
| 1.2.4 Risk-Benefit Assessment | 32 |
| 1.2.5 Potential Risks | 32 |
| 1.2.5.1 Anaphylaxis and Serious Allergic Reactions | 33 |
| 1.2.5.2 Injection Site Reactions | 33 |
| 1.2.5.3 Immune Complex Disease | 34 |
| 1.2.5.4 Infections | 34 |
| 1.2.5.5 Malignancy | 35 |
| 1.2.5.6 Hepatic Function Abnormality | 35 |
| 1.2.5.7 Failure of Vaccination | 36 |
| 1.2.5.8 Potential for Drug-Drug Interactions | 36 |
| 1.2.5.9 Potential Risk to Fetal Development | 36 |
| 2 STUDY OBJECTIVES | 36 |
| 2.1 Phase 1b Multiple Ascending Dose | 36 |
| 2.1.1 Primary Objective | 36 |
| 2.2 Phase 2 Proof of Concept | 37 |
| 2.2.1 Primary Objective | 37 |
| 2.2.2 Secondary Objectives | 37 |
| 3 STUDY ENDPOINTS | 38 |
| 3.1 Phase 1h MAD Study | 38 |

| 3.1.1 | Primary Endpoints | 38 |
|--------|-----------------------------------------------|----|
| 3.1.2 | Exploratory Endpoints | |
| 3.1.3 | Other Endpoints | |
| 3.1.4 | PRO Endpoints. | |
| 3.2 | Phase 2 POC Study | |
| 3.2.1 | Primary Efficacy Endpoint | |
| 3.2.2 | Secondary Efficacy Endpoints | |
| 3.2.3 | Exploratory Endpoints | |
| 3.2.4 | Other Endpoints | |
| 3.2.5 | PRO Endpoints. | |
| 4 S | STUDY PLAN | |
| 4.1 | Study Design | 41 |
| 4.1.1 | Multiple Ascending Dose Phase 1b Study | |
| 4.1.1. | • | |
| 4.1.1. | 2 Dose Limiting Toxicity (DLT) | 42 |
| 4.1.1. | | |
| 4.1.2 | POC Phase 2 Study | 43 |
| 4.1.2. | 1 BOS161721 Dose | 43 |
| 4.1.2. | 2 POC Study Design | 43 |
| 4.2 | Study Schematic | 45 |
| 4.3 | Schedule of Assessments | 46 |
| 5 P | POPULATION | 56 |
| 5.1 | Participant Recruitment | 56 |
| 5.2 | Number of Patients | 56 |
| 5.3 | Patient Screening | 56 |
| 5.4 | Inclusion Criteria | 56 |
| 5.5 | Exclusion Criteria | 58 |
| 5.6 | Concomitant Medications | 60 |
| 5.6.1 | Oral Corticosteroid Dose | 61 |
| 5.6.2 | Other Prohibited and/or Restricted Treatments | 62 |
| 5.7 | Women of Childbearing Potential | 62 |
| 5.7.1 | Determination of Menopause | |
| 5.7.2 | Contraception | 63 |
| 5.8 | Deviation from Inclusion/Exclusion Criteria | 64 |
| 5.8.1 | Patient Withdrawal and Replacement | 64 |
| 5.8.2 | Exception for Non-Responders | 64 |
| 6 S | STUDY PROCEDURES | 65 |
| 6.1 | Screening | 65 |
| 6.1.1 | Retesting During Screening Period | 66 |
| 6.2 | Enrollment/Randomization and Day 1 Treatment | |
| 6.3 | Treatment Period/Follow-Up Visits | 68 |

| 6.4 | Safety Follow-Up Visits | 69 |
|---------|--------------------------------------------------------------|----|
| 6.5 | Premature Discontinuation. | 70 |
| 7 A | SSESSMENTS | 71 |
| 7.1 | Medical History, Demographic and Other Baseline Information | 71 |
| 7.2 | Safety Assessments | |
| 7.2.1 | Laboratory Assessments | |
| 7.2.1.1 | | |
| 7.2.1.2 | | |
| 7.2.2 | Adverse Events | 75 |
| 7.2.2.1 | Definitions | 75 |
| 7.2.2.2 | Recording of Adverse Events | 75 |
| 7.2.2.3 | Severity of Adverse Events | 75 |
| 7.2.2.4 | Causality of Adverse Events | 75 |
| 7.2.2.5 | Seriousness of Adverse Events | 76 |
| 7.2.2.6 | Adverse Events of Special Interest | 77 |
| 7.2.2.7 | Reporting of Adverse Events | 80 |
| 7.2.2.8 | Follow Up of Adverse Events | 82 |
| 7.2.3 | Vital Signs | 82 |
| 7.2.4 | 12-Lead Electrocardiograms | 82 |
| 7.2.5 | Physical Examinations | 83 |
| 7.2.6 | C-SSRS | 83 |
| 7.2.7 | Injection Site Reactions | 83 |
| 7.2.8 | Immunogenicity | 83 |
| 7.3 | Efficacy Assessments. | 84 |
| 7.3.1 | SLEDAI-2K | 84 |
| 7.3.2 | BILAG 2004 | 84 |
| 7.3.3 | PGA of Disease Activity | 84 |
| 7.3.4 | Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response | 85 |
| 7.3.4.1 | SRI-4 Response | 85 |
| 7.3.4.2 | SRI-5 and SRI-6 Response | 85 |
| 7.3.4.3 | BICLA Response | 85 |
| 7.3.5 | CLASI Response | 85 |
| 7.3.6 | ACR-28 Joint Count | 86 |
| 7.3.7 | Laboratory Assessments | 86 |
| 7.4 | Other Variables | 86 |
| 7.4.1 | SLICC/ACR Damage Index | 86 |
| 7.4.2 | PROs | 86 |
| 7.5 | Pharmacokinetic Assessments | |
| 7.6 | Pharmacodynamic Assessments | |
| 7.7 | Pharmacokinetic/Pharmacodynamic Relationship | |
| 7.8 | Protocol Deviations | 87 |

| 8 STUDY DRUG MANAGEMENT | 88 |
|--------------------------------------------------------------|----------|
| 8.1 Description | 88 |
| 8.1.1 Formulation | 88 |
| 8.1.2 Storage | 88 |
| 8.2 Packaging and Shipment | 88 |
| 8.3 Dose and Administration | 88 |
| 8.4 Accountability | 89 |
| 8.5 Prohibited Concomitant Therapy | 89 |
| 8.6 Compliance | 89 |
| 9 STATISTICS | 90 |
| 9.1 Sample Size | 90 |
| 9.2 Statistical Methods | 90 |
| 9.2.1 Analysis Populations | 90 |
| 9.2.2 Demographics and Baseline Characteristics | 91 |
| 9.2.3 Primary Endpoint(s) | 91 |
| 9.2.4 Secondary Endpoint(s) | 91 |
| 9.2.5 Analysis of Safety | 91 |
| 9.2.5.1 Safety Analysis | 91 |
| 9.2.5.2 Data Monitoring Committee | 92 |
| 9.2.6 Pharmacokinetic and Pharmacodynamic Data | 92 |
| 9.2.6.1 Analysis of Pharmacokinetic Data | 92 |
| 9.2.6.2 Analysis of Pharmacodynamic Data | 92 |
| 9.2.6.3 Population Pharmacokinetic Analysis or PK/PD Mod | leling93 |
| 9.3 Interim Analysis and Power | 93 |
| 10 ETHICS AND RESPONSIBILITIES | 94 |
| 10.1 Good Clinical Practice | 94 |
| 10.2 DMC | 94 |
| 10.3 Institutional Review Board/Independent Ethics Committee | |
| 10.4 Informed Consent | 94 |
| 10.5 Records Management | 95 |
| 10.6 Source Documentation | 96 |
| 10.7 Study Files and Record Retention | |
| 11 AUDITING AND MONITORING | 97 |
| 12 AMENDMENTS | |
| 13 STUDY REPORT AND PUBLICATIONS | |
| 14 STUDY DISCONTINUATION | 100 |
| 15 CONFIDENTIALITY | |
| 16 REFERENCES | |
| 17 APPENDICES | |
| APPENDIX 1 NAMES OF STUDY PERSONNEL | |
| APPENDIX 2 DECLARATION OF HELSINKI | 107 |

| APPENDIX 3<br>APPENDIX 4<br>APPENDIX 5 | MEDICATION WASHOUT PERIODS | 112 |
|---|---|---|
| | LIST OF IN-TEXT TABLES | |
| Table 1. | Schedule of Assessments - Phase 1b - Multiple Ascending Dose | 46 |
| Table 2. | Schedule of Assessments - Phase 2 Proof of Concept (POC) Study | 51 |
| Table 3. | Laboratory Tests | 73 |
| Table 4. | Causality Definitions | |
| Table 5. | Sample Size. | |
| | LIST OF IN-TEXT FIGURES | |
| Figure 1. | Individual pSTAT3 C <sub>min</sub> Levels Versus Dose | 31 |
| Figure 2. | Study Diagram for MAD Phase 1b and POC Phase 2 Studies | |
BOS161721 Clinical Study Protocol: BOS161721-02

## LIST OF ABBREVIATIONS

ACR American College of Rheumatology

ADA anti-drug antibody
AE adverse event

AIDS acquired immune deficiency syndrome

ALT alanine aminotransferase
ANA antinuclear antibodies
ANC absolute neutrophil count

APL antiphospholipid

AST aspartate aminotransferase

AUC area under the concentration-time curve

AZA azathioprine

BICLA BILAG-based Composite Lupus Assessment

BILAG British Isles Lupus Assessment Group

BP blood pressure BUN blood urea nitrogen

BW body weight

CD cluster of differentiation

CK creatine kinase C complement

C<sub>L</sub> systematic clearance

CLASI Cutaneous Lupus Erythematosus Area and Severity Index

C<sub>max</sub> maximum plasma concentration

CMH Cochran-Mantel-Haenszel

CS corticosteroids
CSR clinical study report
DILI drug-induced liver injury
DLT dose-limiting toxicity

DMC data monitoring committee

dsDNA double-stranded deoxyribonucleic acid

ECG electrocardiogram
EOT end of treatment

eCRF electronic case report form

F female

Fc fragment crystallizable

FDA Food and Drug Administration FSH follicle stimulating hormone

GCP Good Clinical Practice

eGFR estimated glomerular filtration rate

GLP Good Laboratory Practice

BOS161721

Clinical Study Protocol: BOS161721-02

GWAS genome-wide association studies

γc gamma chain HBV hepatitis B virus

hCG human chorionic gonadotropin

HCl hydrochloride HCV hepatitis C virus

HIV human immunodeficiency virus

HR heart rate

HRT hormone replacement therapy

IA interim analysis

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonization

IEC Independent Ethics Committee

Ig immunoglobulin
IL interleukin

IL-21R interleukin 21 receptor

IM intramuscular INFy interferon gamma

INR International Normalized Ratio IRB Institutional Review Board

IUD intrauterine device

IV intravenous

IVRS interactive voice response system

JAK Janus kinase kg kilogram

KLH keyhole limpet hemocyanin LOCF last observation carried forward

M male

mAb monoclonal antibody
MAD multiple ascending dose

MAPK mitogen-activated protein kinase

MS multiple sclerosis MTX methotrexate

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NIAID/FAAN National Institute of Allergy and Infectious Diseases/Food Allergy and

Anaphylaxis Network

NK natural killer

NOAEL no observed adverse event level

NO nitric oxide

OCS oral corticosteroid

BOS161721 Clinical Study Protocol: BOS161721-02

OTC over-the-counter
PD pharmacodynamics
PEF peak expiratory flow

PGA Physician's Global Assessment

PK pharmacokinetics POC proof of concept

PR (interval) from onset of the p-wave to the end of the r-wave

pSS primary Sjögren's syndrome

pSTAT3 phosphorylated signal transducer and activator of transcription 3

PT preferred term

QRS (interval) from the onset of the q-wave to the end of the s-wave
QT (interval) from onset of the QRS complex to the end of the T wave
QTcF QT interval corrected for heart rate using Fridericia's formula

QFT-G QuantiFERON-TB Gold In-Tube

RA rheumatoid arthritis RNP ribonucleoprotein

RR (interval) from the onset of the r-wave to the onset of the next consecutive r-wave

SAD single ascending dose SAE serious adverse event SAP statistical analysis plan

SC subcutaneous

SDMT safety data monitoring board

CCI

SLE systemic lupus erythematosus SLEDAI-2K SLE Disease Activity Index 2000

SLICC Systemic Lupus International Collaborating Clinics

Sm Smith

SOC system organ class
SRI-4 SLE Responder Index 4
SRI-5 SLE Responder Index 5
SRI-6 SLE Responder Index 6
SSA Sjögren syndrome-A (Ro)
SSB Sjögren syndrome-B (La)

STAT3 signal transducer and activator of transcription 3 SUSAR suspected unexpected serious adverse reaction

 $t_{1/2}$  terminal elimination half-life

TB tuberculosis

TDAR T-cell dependent antibody response

Tfh T-follicular helper

Th T-helper TK toxicokinetics

Clinical Study Protocol: BOS161721-02

T<sub>max</sub> first time to maximum concentration

Treg regulatory T-cell TT tetanus toxoid

ULN upper limit of normal

US United States

Vd volume of distribution

WBC white blood cell

WHO World Health Organization
WOCBP women of childbearing potential

YTE triple mutation

## 1 INTRODUCTION AND RATIONALE

#### 1.1 Indication

BOS161721 is a humanized monoclonal antibody (mAb), which binds to and inhibits interleukin-21 (IL-21) bioactivity, and is being developed for the treatment of moderately to severely active systemic lupus erythematosus (SLE) in adults.

# **1.2** Background and Rationale

#### 1.2.1 Overview of the Disease State

SLE is a chronic inflammatory autoimmune disease that has variable manifestations in multiple organ systems and follows a relapsing and remitting course. The disease process includes abnormal immune responses mediated by tissue-binding autoantibodies and immune complex deposition, giving rise to tissue damage often resulting in end organ disease and even mortality. Survival of SLE has improved due to earlier detection, improved overall medical care, and standardized SLE treatment with corticosteroids, immunosuppressants, and cytotoxic agents. However, some of the morbidity in patients with SLE is related to its treatment. Comparison of early and late outcomes in patients with SLE demonstrate that death in early disease is most commonly due to infections and active SLE causing multi-system organ damage, while thromboses were the most common cause of death during later disease.<sup>2</sup>

The reported prevalence of SLE in the United States (US) is 20 to 70 cases per 100,000 people. More than 90% of cases of SLE occur in women, frequently starting at childbearing age. Women of color are disproportionately affected by SLE. This suggests multiple genetic and environmental factors are at play. Accordingly, a multifactorial view of the immunopathogenesis of SLE suggests more than 1 area of interest, including breach in central tolerance in the adaptive arm of the immune system, peripheral amplification of the autoimmune response by the innate immune system, and local processes in the target organ that facilitate end-organ disease. 4

## **1.2.2 BOS161721 Development**

Boston Pharmaceuticals is developing BOS161721 for the treatment of SLE. BOS161721 is a humanized immunoglobulin G1 (IgG1) mAb directed against human IL-21.

Murine mAb 19E3, the progenitor of BOS161721, was generated using mouse hybridoma technology. 19E3 has subpicomolar (pM) affinity to human IL-21 and was selected for its potent neutralization of IL-21 bioactivity. BOS161721 was generated by the humanization of mAb 19E3 where its complementarity-determining regions were grafted onto a human IgG1 kappa backbone. The fragment crystallizable (Fc) portion of BOS161721 contains a YTE (M252Y/S254T/T256E triple mutation) in the constant domain of the IgG1 heavy chain that was introduced into the parental molecule, 19E3, intended to prolong the in vivo terminal elimination half-life (t<sub>1/2</sub>) of the mAb.<sup>5</sup> Thus, BOS161721 retains sub-pM binding to IL-21 and prevents IL-21 from binding to the IL-21 receptor (IL-21R), inhibiting IL-21 bioactivity.

BOS161721 binds to human IL-21 and Cynomolgus monkey IL-21, which are highly homologous, and neutralizes the bioactivity of both. BOS161721 is specific for IL-21 as it does not bind to or inhibit the other gamma-chain (γc) family of cytokines, and acts to specifically neutralize the IL-21 pathway. In *in vitro* studies, BOS161721 inhibited downstream IL-21-induced signaling, IL-21-induced plasma cell differentiation, and IL-21-induced natural killer (NK) cell activation. In *in vivo* studies, BOS161721 significantly inhibited the T-cell dependent antibody response (TDAR) to immunization with a protein antigen as well as B-cell expansion following a second protein antigen immunization in Cynomolgus monkeys.

#### **1.2.2.1 Interleukin-21**

IL-21 is an inflammatory cytokine, which belongs to a family of cytokines that also includes IL-2, IL-4, IL-7, IL-9, and IL-15, all of which bind to private receptors in complex with the common cytokine receptor yc. Most cytokines in this family are critically important for both the maintenance and function of T-cell and B-cell responses. IL-21 signals through a receptor complex consisting of its own private receptor, the IL-21R and vc. 6,7 Engagement of the IL-21R/γc complex leads to the activation of several signaling pathways, including the Janus kinase/signal transducer and activator of transcription, mitogen-activated protein kinase (MAPK) and phosphoinositide 3-kinase pathways. 8 IL-21 is produced mainly by T-cells and NK T-cells, but neutrophils have also been reported to produce IL-21. 9,10 The IL-21R is expressed on a broad array of cell types, including B-cells, T-cells, NK-cells, macrophages and dendritic cells, as well as other hematopoietic and nonhematopoietic cells such as fibroblasts, keratinocytes, and intestinal epithelial cells. 9,11 Activation of signal transducer and activator of transcription 3 (STAT3) via phosphorylation is critical in regulating human B-cell responses to IL-21<sup>12</sup>; phosphorylated STAT3 (pSTAT3) forms a homodimer, which translocates to the nucleus where it initiates transcription of the IL-21 gene, forming an autocrine loop for IL-21 production via STAT3 phosphorylation. <sup>13</sup> In addition, IL-21 has been shown to upregulate expression of its own receptor <sup>14</sup> and induces an autocrine feedback loop. <sup>15</sup>

IL-21 modulates various aspects of immune function. It promotes cluster of differentiation 4 (CD4+) T-cell differentiation and promotes the generation of T-helper (Th)17<sup>16</sup> and T-follicular helper (Tfh) cells. <sup>15,17</sup> In mice, IL-21 has been shown to regulate the balance between Th17 and regulatory T-cell (Treg), in that it increases Th17, while inhibiting Treg differentiation. <sup>18</sup> Less is understood with regards to human Tregs, although IL-21 has been reported to counteract Treg suppression of human effector T-cells and blockade of IL-21 promotes Treg generation in a murine model of graft versus host disease induced by human T-cells. <sup>20</sup> IL-21 upregulates CD8+ T-cell and NK-cell expansion and cytolytic activity by increasing granzyme B and perforin. <sup>21,22</sup> IL-21 also has been reported to increase granzyme B in plasmacytoid dendritic cells and B-cells resulting in inhibition of T-cell responses. <sup>23,24</sup> IL-21 also has a variety of effects on nonhematopoietic cells, such as stromal cells and induces inflammation through matrix metalloproteinase release by gut intestinal fibroblasts. <sup>25</sup>

One principal non-redundant role of IL-21 is the promotion of B-cell activation, differentiation, or death during humoral immune responses. <sup>14</sup> Furthermore, increased IL-21 production is characteristic of several autoimmune diseases and is likely to contribute to autoantibody production as well as pathologic features of autoimmune disease. <sup>26</sup> The critical role of IL-21 in promoting humoral and other immune responses makes it an important focus of potential

therapeutic interventions in conditions characterized by overproduction of pathogenic autoantibodies. IL-21 production by Tfh cells in humans is believed to play a major role in driving the autoantibody production through its role in plasma cell differentiation. Importantly, Tfh cell populations are expanded in patients with autoimmune diseases such as lupus, bullous pemphigoid, rheumatoid arthritis (RA) and primary Sjögren's syndrome (pSS) and have been reported to correlate with IL-21 levels, autoantibodies, and disease severity. <sup>26,27,28,29</sup> Furthermore, loss of number and functionality of Tregs has been associated with autoimmune diseases such as SLE and giant cell arteritis, which IL-21 is expected to modulate. <sup>30,31</sup> Thus, neutralization of IL-21 in settings of autoimmunity is expected to impact several cell populations believed to be involved in the pathogenesis of autoimmune disorders including SLE.

BOS161721 selectively binds IL-21 with high affinity to neutralize IL-21, and due to its pleiotropic nature, neutralization of IL-21 is expected to impact several cell populations believed to be involved in the pathogenesis of SLE. Importantly, patients with SLE have elevated IL-21 plasma levels that correlate with the severity of the disease. Recently, genome-wide association studies (GWAS) have provided convincing evidence that the chromosomal 4q 27 region harbors the IL-21 genes and is associated with chronic inflammatory disorders, including SLE.<sup>29</sup>

#### 1.2.2.2 Preclinical Studies

The pharmacokinetics (PK) of BOS161721 were characterized following single-dose intravenous (IV) administration of BOS161721 (0.01 to 30 mg/kg) in male Cynomolgus monkeys or repeat, every 2 weeks IV administration (15 to 100 mg/kg) and subcutaneous (SC) administration (50 mg/kg) in male and female Cynomolgus monkeys. Systemic exposure was approximately dose-proportional within the tested dose range. SC bioavailability was determined to be 64.3%.

Two single-dose (IV) non-good laboratory practice (GLP) studies conducted in Cynomolgus monkeys evaluated the toxicity, pharmacodynamics (PD), toxicokinetics (TK), and immunogenicity of BOS161721. Following a single IV administration (slow bolus), there were no BOS161721-related adverse changes, resulting in a no-observed-adverse-effect-level (NOAEL) value of 30 mg/kg, the highest dose tested among 2 studies.

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) administration for 3 months (a total of 7 doses).



#### 1.2.2.3 Clinical Studies

BOS161721-01 was a double-blind, Phase 1, single ascending dose (SAD) study to assess the safety, PK, and PD of BOS161721 in healthy subjects. The primary objective of the study was to characterize the safety and tolerability of IV and SC SADs of BOS161721 in an otherwise healthy subject population without concomitant illnesses, immune abnormalities, or concomitant medications. Secondary objectives included characterization of the PK and immunogenicity of BOS161721, and exploratory objectives included the evaluation of the effect of BOS161721 on TDAR to keyhole limpet hemocyanin (KLH) (primary and secondary immunizations) in healthy subjects, the effects of BOS161721 on plasma levels of IL-21 (free and bound), and the evaluation of the effect of BOS161721 on IL-21 gene expression (via gene signature) in blood. This study consisted of 8 cohorts. Subjects were randomized in a 3:1 ratio (BOS161721: placebo) and received either a single dose of BOS161721 (1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg) or placebo, with safety follow-up. For the first cohort, after the first 2 subjects were dosed (1 active and 1 placebo), there was a minimum gap of 48 hours before the remaining subjects from that cohort were dosed, to allow for an initial review of any emerging safety and tolerability data. For all cohorts, escalation to the next dose was not sooner than 8 days after all the subjects in the prior cohort had been dosed and were based on a review of at least 7 days of safety and tolerability data by the Safety Data Monitoring Team (SDMT).

Blood samples were collected at every in-house study visit for BOS161721 concentration determinations. Blood samples were also collected for determination of IL-21 plasma levels (free and total). Safety was assessed based on the occurrence of treatment-emergent AEs, hepatic function abnormality, and acute and delayed hypersensitivity reactions. Other safety variables included electrocardiograms (ECGs), vital signs (blood pressure, heart rate, and temperature), safety laboratory assessments, blood sampling for ADAs, total IgG and IgM levels, CD4+ count, and full and targeted physical examinations. Overall, there were no clinically significant findings from this study; there were no serious adverse events (SAEs), deaths, or discontinuations due to AEs during the study, AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs. PK data from the SAD study demonstrates BOS161721 has an extended t<sub>1/2</sub> (provisional single dose data indicates this to be approximately 42-46 days) which supports evaluation of monthly dosing.

# 1.2.3 Study Dose Selection

Doses have been selected for the multiple ascending dose (MAD) Phase 1 study based on a 90-day safety, tolerability, PK, and PD data review from the Phase 1 SAD study (BOS161721-01); the SDMT reviewed the blinded safety data from subjects for each dose cohort (8 cohorts, evaluating 1 [IV], 3 [SC], 10 [SC], 22 [IV], 30 [SC], 60 [SC], 120 [SC], or 240 [SC] mg), along with the accumulated safety and available PK/PD data from all subjects in the previous dose cohorts, to make a decision on whether to proceed to the next higher dose level, repeat a dose level, or stop dose escalation. Overall, there were no clinically significant safety or tolerability findings from this study.

Based on the Day-90 interim cut of the PK and biomarker data in the BOS161721-01 study, the recommended doses for evaluation in the MAD phase of this study are 20, 60, and 120 mg SC monthly. This dose recommendation is supported by evidence of linear PK with BOS161721 resulting in a median T<sub>max</sub> of 6 days and an apparent terminal half-life of 44 days. Furthermore, pSTAT3 suppression, a marker of IL-21 target engagement, follows a similar time course of the mAb levels, with maximal and sustained suppression apparent with doses greater than 30 mg SC (Figure 1).



Figure 1. Individual pSTAT3 C<sub>min</sub> Levels Versus Dose

IV = intravenous, pSTAT3 = phosphorylated signal transducer and activator of transcription 3; SC = subcutaneous

All doses selected for the MAD study are projected not to exceed peak levels or exposure of that achieved following the highest single dose of 240 mg SC administered in the Phase 1 SAD study. Cohort 1 will include randomized treatment to the 20 mg dose. Based on the staggered study design, the data monitoring committee (DMC) will perform a scheduled review of safety data and sequentially consider dose escalation for Cohorts 2 and 3. In addition, the DMC will conduct a data review for the first interim analysis (IA1) to determine which dose will be carried forward into the proof of concept (POC) Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 from the MAD study (see Section 4.1.1.1).

#### 1.2.4 Risk-Benefit Assessment

The available preclinical data on BOS161721, the findings in clinical study BOS161721-01, and existing clinical information on IL-21 inhibitors suggest that the present clinical study has an acceptable risk-benefit ratio. In this study, the risk-benefit assessment of BOS161721 in adult patients with moderately to severely active SLE will be ongoing, with step-wise evaluations during the staggered MAD study. The DMC used in this study is charged with assessing such actions in light of an acceptable benefit-risk profile for BOS161721 as an anti-IL-21 mAb. Formal DMC monitoring meetings will occur as described in the DMC Charter. Two weeks after Cohort 1 has received a second dose of study drug, the DMC will evaluate the safety and tolerability data from Cohort 1 to determine the recommended dose for Cohort 2. Two weeks after 8 patients in Cohort 2 receive a second dose, the DMC will determine if dose escalation to Cohort 3 can proceed. Two weeks after the last patient in Cohort 3 receives the second dose, the DMC will conduct a data review for the IA1 to determine which dose will be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2 and 3 during the MAD study. Thereafter, DMC monitoring will be conducted periodically throughout the study as described in the DMC charter. With the agreement of the DMC and sponsor, this schedule may be modified depending on the rate of patient accrual. Additional details can be found in the DMC Charter.

The benefit of participation for all patients in this study is close monitoring of their medical condition and safety of their treatment. Those randomized to the active treatment arm may potentially experience improvement in their SLE disease. Those randomized to the placebo (in combination with standard of care) arm are not expected to obtain any additional benefit, beyond those of their background treatment, though close monitoring of their medical condition and safety may itself be associated with improving their SLE.

#### 1.2.5 Potential Risks

Potential risks based on the mechanism of action of BOS161721 include infections, risks associated with the administration of any foreign protein or biologic agent, including injection site reaction, anaphylaxis, serious allergic reaction, and development of ADAs. ADAs could result in immune complex disease (with manifestations such as arthralgias, serum-sickness, and vasculitis), autoimmunity, or altered BOS161721 levels or activity. Further details can be found

in the current Investigator's Brochure (IB) for BOS161721, which contains comprehensive toxicology, preclinical and clinical information on BOS161721.

Two investigational drug products are considered to be in the same pharmacological class as BOS161721 based on interruption of signaling through the IL-21 signaling pathway. No potential risk generalizable across the class has been observed with these investigational products. Based on the clinical Phase 1 SAD study (BOS161721-01), AEs reported as related to the study drug, particularly infections (flu-like symptoms, etc), were expected for the compound, and there were no clinically relevant changes in laboratory and ECG results or vital signs.

The majority of IgG elimination occurs via intracellular catabolism, following fluid-phase or receptor-mediated endocytosis. This type of endocytosis and elimination is a form of target-mediated disposition where the interaction of the drug and its pharmacological target (eg, a target receptor) serves as a significant contributor to the kinetics of antibody distribution and elimination. Renal elimination, which is a primary pathway of clearance of small-molecule drugs, is relatively unimportant for IgG, as its large size prevents efficient filtration through the glomerulus. Secretion into the bile is an important pathway of elimination of IgA antibodies, but this route is not a significant contributor to the elimination of IgG antibodies. Thus, risk to renal and hepatic systems due to metabolism of BOS161721 is low.<sup>33</sup>

# 1.2.5.1 Anaphylaxis and Serious Allergic Reactions

As with the administration of any foreign protein and/or other biological agents, acute hypersensitivity reactions, including acute anaphylactic/hypersensitivity, severe allergic, and anaphylactoid reactions may follow infusion of mAbs and can be caused by various mechanisms. These acute hypersensitivity reactions may be severe and result in death.

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria,<sup>34</sup> and are discussed in Section 7.2.2.6.1.

Based on the limited Phase 1 SAD study (BOS161721-01), anaphylaxis and serious allergic reactions in subjects who received BOS161721 was not observed.

Patients with a known history of allergy or severe hypersensitivity reaction to any component of BOS161721 formulation or patients with a history of anaphylaxis to any other biological therapy such as mAbs will be excluded from studies with BOS161721. In addition, appropriate drugs and medical equipment to treat acute hypotensive, bronchoconstrictive, or anaphylactic reactions will be immediately available at the unit and study personnel will be trained to recognize and treat these reactions.

## 1.2.5.2 Injection Site Reactions

In a repeat-dose GLP toxicology study in Cynomolgus monkeys, BOS161721 was administered every 2 weeks by IV or SC (50 mg/kg) for 3 months (a total of 7 doses); no SC animals had injection reactions.

Based on the Phase 1 SAD study (BOS161721-01), incidence of injection site reactions in subjects who received BOS161721 was similar to placebo.

Patients will be monitored for local injection site reactions in this study. See Section 7.2.7.

# **1.2.5.3 Immune Complex Disease**

The potential risk of immune complex disease for BOS161721 is theoretical, based on the known risks associated with mAbs. The administration of a mAb can result in the formation of ADAs. Administration of the mAb in the presence of ADA may result in the formation of circulating antibody-antigen complexes potentially resulting in altered BOS161721 levels or activity or deposition of the complexes in microvasculature. Complement is frequently involved in the latter setting, and the breakdown products of complement attract polymorphonuclear leukocytes to the site of deposition where they can provoke local tissue damage through specific or nonspecific release of enzymes. Two of the more common end-organ targets are the blood vessels (vasculitis) and kidney (nephritis). These clinical manifestations represent immune complex disease or Type III hypersensitivity. Although BOS161721 is a humanized mAb, ADAs may develop; however, the likelihood of occurrence of immune complex disease with BOS161721 is low. The findings of immune complex disease are typically reversible when mAb administration stops and the antibody-antigen complexes are cleared from the body.

Based on the limited Phase 1 SAD study (BOS161721-01), immune complex disease in subjects who received BOS161721 was not observed.

## 1.2.5.4 Infections

BOS161721 is expected to diminish the activity of T-cell, B-cell and NK-cell lines. Like other medications modulating immune response, BOS161721 may increase the potential risk for infection, including serious infections. IL-21 produced by CD4+ Th cells is required to sustain the anti-viral function of CD8+ T-cells against chronic viral infections. Nonclinical evidence suggests that the risk of chronic viral infection recurrence or increased severity may occur with IL-21 inhibition.<sup>35</sup>

These conditions will be fully characterized with clinical descriptions and routine laboratory and/or specialty testing and treated where indicated with appropriate local standard of care.

Patients with a history of opportunistic infection, including recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years, or any other underlying pathology predisposing to serious infection, are excluded from studies with BOS161721 (for further details please refer to the current IB for BOS161721).

Patients will be assessed for hepatitis B, and C, and HIV-1/2 combination, at screening.

# Cryptosporidium Infection

Cryptosporidium infection was noted in patients with an IL-21 receptor loss-of-function gene mutation and similar findings of cryptosporidium infection have been observed in immunosuppressed liver transplant and human immunodeficiency virus patients. <sup>36,37</sup> Since

BOS161721 is expected to diminish the immunosurveillance activity of T-cell, B-cell, and NK-cell lines, a similar risk is biologically plausible with prolonged exposure to BOS161721.

Since the risk of opportunistic cryptosporidium infection increases with low levels of CD4+ T-cells, <sup>37</sup> patients with a CD4+ count < 500 cell/mm<sup>3</sup> were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from the proposed MAD/POC studies. Patients exposed to investigational product who develop diarrhea during the course of the study should immediately undergo an assessment for opportunistic infection including stool for ova and parasites and stool examination for cryptosporidium. Positive cryptosporidium in stool sample at screening is an exclusion. Treatment by the investigator where indicated should be guided by findings and be consistent with local standard of care.

Based on the limited Phase 1 SAD study (BOS161721-01), infections in subjects who received BOS161721 was not observed.

# 1.2.5.5 Malignancy

The stimulatory effect of IL-21 on NK cells and CD8+ T-cells suggests the cytokine may have anti-tumor activity. Nonclinical studies have demonstrated significant anti-tumor effects of IL-21 in a number of tumor models. IL-21 therapy of human metastatic melanoma and renal cell carcinoma has demonstrated POC with significant increases in levels of perforin, granzyme B, and interferon gamma (IFN $\gamma$ ) expression in CD8+ T-cells and NK T-cells. Clinical response has been limited in these generally unmanageable diseases.

The impact of treatment with anti-IL-21 therapy on the development or growth of malignancies is not known; however, as with other immunomodulatory biologic agents, treatment with BOS161721 may result in an increase in the risk of malignancies. NK cell suppression by IL-21 neutralization may represent a biological mechanism for a potential risk for malignancy. Patients with a history or current diagnosis of cancer within the past 5 years, with the exception of non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy, are excluded from the study.

Based on the limited Phase 1 SAD study (BOS161721-01), malignancy in subjects who received BOS161721 was not observed.

## **1.2.5.6** Hepatic Function Abnormality

There is no substantial evidence suggesting BOS161721 is associated with liver function abnormality. However as a precaution, patients with a history of abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), or bilirubin at screening (ALT/AST >  $2 \times \text{upper limit of normal [ULN]}$ ; total bilirubin >  $1.5 \times \text{[ULN]}$  and judged by the investigator to be clinically significant) were excluded from the Phase 1 SAD study (BOS161721-01), and will be excluded from the MAD study. Patients with a positive hepatitis B or C test or a history of alcohol dependence will also be excluded.

Based on the limited Phase 1 SAD study (BOS161721-01), hepatic function abnormality in subjects who received BOS161721 was not observed.

#### 1.2.5.7 Failure of Vaccination

IL-21 is a key cytokine in development of B-cells into immunoglobulin-secreting plasma cells. Abnormal signaling through the IL-21R/Janus Kinase (JAK)3/signal transducer and activator of transcription (STAT3) pathway leads to defective humoral immune responses to both T-dependent and T-independent antigens and impairs the establishment of long-lasting B-cell memory. Abnormal signaling through the pathway has been related to decreased specific antibody responses following vaccination, and to increased susceptibility to encapsulated bacterial infections.<sup>38</sup>

The effect of BOS161721 was evaluated in in vivo single dose studies in Cynomolgus monkey in which the animals received vaccination to T-cell dependent KLH antigen to stimulate a TDAR. These in vivo studies demonstrated that BOS161721 significantly inhibited B-cell proliferation and IgG antibody responses to the KLH protein antigen; however, it is worth noting that BOS161721 administration did not produce any remarkable changes in anti-KLH antibody data for IgM, IgG1, IgG3, and IgG4 or anti-tetanus toxoid (TT) antibody data for IgM, IgG, IgG1, or IgE during the dosing phase in the same study.

## 1.2.5.8 Potential for Drug-Drug Interactions

Drug-drug interactions were not evaluated in the Phase 1 SAD study (BOS161721-01), which included only healthy adult subjects. Use of prescription medications (with the exceptions of oral contraceptives), and over-the-counter (OTC) treatments including herbal supplements such as St John's Wort (except multivitamins), in the 2 weeks prior to screening was prohibited in the SAD study.

See Section 5.5 for other specific exclusion criteria which support lowered risk of interactions, and Section 5.6.1 for corticosteroid (CS) dosing. In addition, Section 1.2.5.6 describes considerations for hepatic function for this study.

## 1.2.5.9 Potential Risk to Fetal Development

No data on preclinical reproductive toxicity are available at the time of this study.

#### 2 STUDY OBJECTIVES

This trial has separate primary and secondary objectives for the MAD Phase 1b and POC Phase 2 studies.

# 2.1 Phase 1b Multiple Ascending Dose

# 2.1.1 Primary Objective

To assess safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20 mg, 60 mg, and 120 mg) administered SC in adult patients with moderately to severely active SLE on limited background standard of care treatment, in order to estimate the optimal dose.

BOS161721 Clinical Study Protocol: BOS161721-02

# 2.2 Phase 2 Proof of Concept

# 2.2.1 Primary Objective

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on the SLE Responder Index 4 (SRI-4), with sustained reduction of oral CS, in adult patients with moderately to severely active SLE on limited background standard of care treatment.

## 2.2.2 Secondary Objectives

To demonstrate a superior effect of BOS161721 at the chosen dose compared with placebo for response on clinical indicators of SLE activity, in adult patients with moderately to severely active SLE on limited background standard of care treatment, including:

- Changes in SLE-specific autoantibody titers;
- Changes in complement 3 and 4 (C3 and C4) levels;
- Responses on SRI-4, SRI-5, and SRI-6, with sustained reduction of oral CS;
- Response on the British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (BICLA);
- Response on the Cutaneous Lupus Erythematosus Area and Severity Index (CLASI);
- Changes in the SLEDAI-2K;
- Changes in American College of Rheumatology (ACR)-28 joint count.

## 3 STUDY ENDPOINTS

This trial has separate primary and secondary endpoints for the MAD Phase 1b and POC Phase 2 studies.

# 3.1 Phase 1b MAD Study

# 3.1.1 Primary Endpoints

Evaluation of safety, tolerability, and immunogenicity at each dose level, to determine the optimal dose, will include the recording of the following parameters:

- Incidence and severity of AEs, AEs of special interest, and SAEs;
- 12-lead ECGs;
- Vital signs (blood pressure [BP], heart rate, and temperature);
- Clinical laboratory assessments;
- Physical examinations;
- Evaluation for ADAs.

# 3.1.2 Exploratory Endpoints





# 3.2 Phase 2 POC Study

# 3.2.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the proportion of patients who achieve treatment response as measured by the SRI-4 at Week 28, along with a sustained reduction of oral CS ( $\leq$  10 mg/day and  $\leq$  Day 1 dose) between Week 16 and Week 28.

## 3.2.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints are:

- The proportion of patients who achieve treatment response for the SRI-5 and SRI-6 at Week 28, along with a sustained reduction of oral CS (≤ 10 mg/day and ≤ Day 1 dose) between Week 16 and Week 28;
- Changes from baseline in dsDNA, ANA, SSA, SSB, RNP, Sm, APL autoantibodies, at Week 16 and Week 28;
- Changes from baseline in C3 and C4 levels at Week 16 and Week 28;
- Changes from baseline in the SLEDAI-2K at Week 28;

- Time to BILAG A or B flare;
- Changes from baseline in the CLASI at Week 28;
- The proportion of patients with a BICLA response at Week 28;
- The proportion of patients with CLASI response at Week 28;
- Changes from baseline (percentage) in swollen joints and tender joints ACR-28 joint count;
- Incidence and severity of AEs, AEs of special interest, and SAEs;
- 12-lead ECGs;
- Vital signs (BP, heart rate, and temperature);
- Clinical laboratory assessments;
- Physical examinations and targeted physical examinations;
- Evaluation for ADAs.

# 3.2.3 Exploratory Endpoints

• CCI
• CCI
• CCI
• CCI
• CCI
• CCI

# 3.2.4 Other Endpoints

• CCI

| • | CCI | |
|-----|-----|---------------|
| • | CCI | |
| 3.2 | .5 | PRO Endpoints |
| • | CCI | |

#### 4 STUDY PLAN

# 4.1 Study Design

This is a Phase 1b/2 combined, randomized, multicenter, double-blind, placebo-controlled trial to study the clinical efficacy, safety, and PK of SC doses of BOS161721 in adult patients with moderately to severely active SLE. After successfully completing a screening phase, patients will be randomized to a specified dose of BOS161721 or placebo. The dosing schedule will be monthly.

The trial will consist of 2 studies: MAD Phase 1b, and POC Phase 2. Both studies will be double-blinded, and patients will have the same number of visits. Patients may receive a total of 7 SC monthly doses of study drug on Days 1, 30, 60, 90, 120, 150, and 180, followed by a 90-day safety follow-up visit.

SLE disease activity assessment data will be centrally reviewed by medical monitor and sponsor to ensure the scores are clinically meaningful and compliant with specific definition. The scope of responsibility includes, but is not limited to, review and confirmation of "A" and "B" BILAG system organ disease, confirmation of clinical components of the SLEDAI-2K score at screening and during the study, and cross-validation of the instruments used in this study to assess the disease being studied. Further details on the content and methods of data reports by the medical monitor and sponsor will be outlined in the Medical Data Review Plan along with the processes and procedures that will be followed.

## 4.1.1 Multiple Ascending Dose Phase 1b Study

The MAD study will consist of 3 cohorts:

- Cohort 1 (20 mg SC) will include 6 patients
  - o 5 patients will receive BOS161721 (active group) and 1 patient will receive placebo (placebo group)

BOS161721 Clinical Study Protocol: BOS161721-02

- Cohorts 2 (60 mg SC) and 3 (120 mg SC) will include 12 patients each
  - o 9 patients in the active group and 3 in the placebo group

Doses selected for each of the 3 cohorts is based on a 90-day safety, tolerability, PK and PD data review from the Phase 1 SAD study (BOS161721-01) in healthy subjects. All doses selected for the MAD study are projected not to exceed the mean peak levels or exposures of that achieved in the SAD study.

#### **4.1.1.1 Dose Escalation for the MAD Study**

The MAD study design is staggered, where after the 6 patients in Cohort 1 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 2 begins dosing (after DMC evaluation of the safety and tolerability data from Cohort 1). Similarly, after 8 of the 12 patients in Cohort 2 have received 2 doses and have completed 2 weeks of follow-up after the second dose, Cohort 3 begins dosing (based on the dose level determined after DMC evaluation of the safety and tolerability data from Cohorts 1 and 2). Two weeks after the last patient in Cohort 3 receives the second dose, the DMC will conduct a data review for the IA1 to determine which dose will be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available when the last patient in Cohort 3 reaches 60 days (dose 2). Each cohort will continue at their assigned dose level through their respective 6-month treatment periods (See Study Schematic, Section 4.1). If > 3 patients discontinue the study in a cohort, he/she will be replaced.

Criteria for dose escalation are further described in the DMC Charter. See Section 4.1.1.2 for additional details about DLTs.

## **4.1.1.2 Dose Limiting Toxicity (DLT)**

Severity of adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs occurring after study drug administration, which are attributable to the study drug, will be considered DLTs:

# **Hematologic:**

- Grade 4 neutropenia;
- Grade 3 neutropenic infection;
- Grade 3 thrombocytopenia with bleeding;
- Grade 4 thrombocytopenia.

#### **Non-Hematologic:**

• Grade 3 or above toxicities, persisting after optimal treatment with standard medical therapy (eg, anti-emetics, anti-diarrheals);

• Drug-induced liver injury ([DILI], Hy's Law), as defined in Section 7.2.2.6.3.

Investigators should always manage their patients according to their medical judgment which may include interruption of study drug based on the particular clinical circumstances. All dose modifications/adjustments must be clearly documented in the patient's source notes and electronic Case Report Form (eCRF).

#### 4.1.1.3 DMC Recommendations

During scheduled meetings, the DMC will review relevant study data for safety or benefit-risk concern. During the MAD study, the DMC may provide the following recommendations to the sponsor:

- Expanding a cohort at a specific dosing level, or repeating a lower dose in a subsequent cohort:
- Continuing a dose level for a given cohort;
- Escalating a dose level for a subsequent cohort;
- Termination of current or previous cohort(s).

Further dosing in a given cohort will be halted if 2 or more DLTs are identified intra- and inter-patients dosed. For the POC study, the DMC will conduct a data review for the IA1 to determine which dose will be carried forward into the POC Phase 2 study. This POC dose decision will be based on evaluation of the PK, safety (inclusive of dose-limiting toxicity [DLT]), and tolerability data (and available PD/biomarker data) from Cohorts 1, 2, and 3; this dose will not exceed doses tested during the MAD study. The DMC will be reviewing all relevant data from Cohorts 1, 2, and 3 that is available when the last patient in Cohort 3 reaches 60 days (dose 2). Details are provided in the DMC Charter.

# 4.1.2 POC Phase 2 Study

#### 4.1.2.1 BOS161721 Dose

The optimal dose evaluation is chosen based on MAD Phase 1b safety results. The dose will be communicated by a letter to site investigators participating in the POC Phase 2 study, and to the IRB/IEC. Once the POC dose decision has been made, screening for the POC study can begin.

## 4.1.2.2 POC Study Design

For the POC study, 156 patients will be randomized to active or placebo groups in a 2:1 ratio.

BOS161721 Clinical Study Protocol: BOS161721-02

As in the MAD study, each patient in the POC study may receive a total of 7 SC monthly doses of study drug on Days 1, 30, 60, 90, 120, 150, and 180. Assessments will be completed according to the Schedule of Assessments (Section 4.3). Dose selection will be based on the sponsor's assessment of safety, tolerability, immunogenicity, and PK and PD data from the MAD study of 30 patients treated with BOS161721/placebo.

Data from approximately 60 patients (including the 12 from the MAD study, or 6 fewer if the low dose is chosen who are in the cohort of the chosen dose for the POC study) who complete 3 months of treatment will be used in the IA2 at Week 16 to assess if the trial could stop for an early futility conclusion (see Section 9.3 for details regarding the IA). If futility is not claimed in the IA2, the POC study will continue to 156 patients.

Following the 6-month treatment period, primary and secondary efficacy endpoints will be assessed for each patient after providing their 24-week disease activity assessments.

DMC monitoring will be conducted periodically throughout the study as described in the DMC charter.

BOS161721 Boston Pharmaceuticals, Inc. Clinical Study Protocol: BOS161721-02

# 4.2 Study Schematic

Figure 2. Study Diagram for MAD Phase 1b and POC Phase 2 Studies



A = active drug (BOS161721); P = placebo


Clinical Study Protocol: BOS161721-02

# 4.3 Schedule of Assessments

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | | Tro | eatment | Period | Follow- | Up | | | | F | Safety<br>ollow-U | p |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | | | 7 | 8 | 9 |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | | | |
| Serum pregnancy test (women) | X | | | | | | | | | | | | | | | |
| FSH and estradiol<br>(postmenopausal<br>women) | X | | | | | | | | | | | | | | | |
| TB test<br>(QuantiFERON-TB<br>Gold In-Tube) <sup>b</sup> | X | | | | | | | | | | | | | | | |
| Chest x-ray <sup>b</sup> | X | | | | | | | | | | | | | | | |
| Serology (hepatitis B and C, HIV-1/2 combination) | X | | | | | | | | | | | | | | | |
| SLICC Criteria for<br>SLE | X | | | | | | | | | | | | | | | |
| Stool sample <sup>c</sup> | X | | | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | | | X | | | X | | | | | |
| Randomization <sup>d</sup> | | X | | | | | | | _ | | | | | | | |


Clinical Study Protocol: BOS161721-02

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | | Tre | eatment | Period | Follow- | Up | | | | F | Safety<br>ollow-U | р |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | | | 7 | 8 | 9 |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| General | | | | | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | | X | | X | X | X | X | X | | | | | |
| Injection site reaction assessment <sup>e</sup> | | X | | | X | | X | X | X | X | X | | | X | X | X |
| Targeted physical examination | | | | X | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>f</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| Urine pregnancy test (women) <sup>g</sup> | | X | | | X | | X | X | X | X | X | | | | | |
| Spot urine for protein/creatinine | | | | | ** | | | *** | 7.7 | | 77 | | | *** | | *** |
| ratio | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Concomitant medication <sup>h</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| AEs and SAEs | | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| BILAG-2004 Index | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLEDAI-2K | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| PGA of disease activity | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLICC/ACR Damage | | X | | | | | | | | | X | | | | | |


Clinical Study Protocol: BOS161721-02

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | | Tre | eatment | Period | Follow- | ·Up | | | | F | Safety<br>ollow-U | р |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | | | 7 | 8 | 9 |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| Index | | | | | | | | | | | | | | | | |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| 12-lead ECG <sup>i</sup> | X | X | | | X | | | X | | | | | | | | X |
| Laboratory | | | | | | | | | | | | | | | | <u> </u> |
| CD4+ count | X | X | | X | X | X | | X | | | X | | | | | _ |
| Clinical laboratory<br>assessments<br>(hematology and | | | | | | | | | | | | | | : | | |
| clinical chemistry) | X <sup>j</sup> | X | | | X | X | X | X | X | X | X | | | X <sup>j</sup> | X | X |
| Coomb's test direct <sup>k</sup> | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | | X | X | X | | X | | | X | | | | | <u> </u> |
| Plasma CC | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Plasma CCI & | X | X | | X | X | | X | X | | | X | | | | | |
| Whole blood for leukocyte immunophenotype | X | X | | X | X | | X | X | | | X | | | | | |
| ADA | | X | | X | X | | X | X | | | X | | | | | X |
| nAb <sup>m</sup> | | | | | | | | X | | | X | | | | | |
| pSTAT3 | | X | | | X | X | X | X | | | X | | | | | X |
| CCI | | X | | | | | | | | | X | | | | | |
| Whole blood RNA collection | | X | | X | X | | | X | | | | | | | | X |
| CCI | X | X | | | X | | X | X | X | X | X | | | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> |


Clinical Study Protocol: BOS161721-02

Table 1. **Schedule of Assessments - Phase 1b - Multiple Ascending Dose** 

| | Screen <sup>a</sup> | Enroll | | | | Tro | atment | Period | Follow- | Up | | | | F | Safety<br>ollow-U | р |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | 1.5 | 2 | | 7 | 8 | 9 | | | | | |
| Weeks | | | 1 | 2 | 4 | 6 | 26 | 28 | 32 | 36 | | | | | | |
| Dane | -28 | 1 | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | $(\pm 3)$ | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| CRP | X | | | | | | | X | | | | | | | | X |
| PK Labs | | | | | | | | | | | | | | | | |
| Predose <sup>o</sup> | | X | | | X | | X | X | X | X | X | | | | | |
| Postdose | | X <sup>p</sup> | X | X | X <sup>p</sup> | | | | | | X <sup>p</sup> | X | X | X | X | X |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index;

CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram;

; FSH = follicle stimulating hormone; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G;

IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; nAb = neutralizing antibody; PGA = Physician's Global Assessment;

PK = pharmacokinetic; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; RNA = ribonucleic acid; RNP = ribonucleoprotein;

SAE = serious adverse event; SC = subcutaneous; CC ; SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; CC

Screening assessments will be performed over more than 1 visit.

TB = tuberculosis; TDAR = T-cell dependent antigen response.

- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 1).
- Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- Randomization should occur after patient eligibility has been confirmed by central eligibility review.
- Injection site reaction assessments to be performed predose and at 2 hours postdose.
- Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 1 at predose and at 1 and 2 hours postdose as well as on each of the scheduled outpatient days in the table above. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.
- Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 1 (randomization day). See Section 5.6.1 for further details.
- ECG will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws.


Clinical Study Protocol: BOS161721-02

 Table 1.
 Schedule of Assessments - Phase 1b - Multiple Ascending Dose

| | Screen <sup>a</sup> | Enroll | | | | Tre | atment | Period | Follow- | Up | | | | F | Safety<br>ollow-U | p |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | 1.5 | | 7 | 8 | 9 | | | | | | |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| | -28 | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ | (± 3) | $(\pm 3)$ |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |

Clinical laboratory assessments will include a fasting glucose and lipid panel during screening and Week 28.


When clinically indicated.

Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.

m nAb is assessed if patient is positive for ADA.

<sup>&</sup>lt;sup>n</sup> Only dsDNA collected during safety follow-up visits.

OPPREDOR Predose samples occur on study drug administration visit days.

Postdose samples will be collected at 4, 8, and 24 hours after study drug administration on Days 1, 30, and 180.

Clinical Study Protocol: BOS161721-02

 Table 2.
 Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screen <sup>a</sup> | Enroll | | | | 7 | [reatme | nt Perio | d Follow | -up | | | | Safet | y Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | | | 7 | 8 | 9 |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| _ | | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | -28 to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| Full physical exam | X | X | | | | | | | | | | | | | | |
| Serum pregnancy<br>test (women) | X | | | | | | | | | | | | | | | |
| FSH and estradiol<br>(postmenopausal<br>women) | X | | | | | | | | | | | | | | | |
| TB test<br>(QuantiFERON-TB<br>Gold In-Tube) <sup>b</sup> | X | | | | | | | | | | | | | | | |
| Chest x-ray <sup>b</sup> | X | | | | | | | | | | | | | | | |
| Serology (Hepatitis<br>B and C; HIV-1/2<br>combination) | X | | | | | | | | | | | | | | | |
| SLICC Criteria for<br>SLE | X | | | _ | | | | | | | | _ | _ | | | |
| Stool sample <sup>c</sup> | X | | | | | | | | | | | | | | | |
| C-SSRS | X | X | | | | | | X | | | X | | | | | |
| Randomization <sup>d</sup> | | X | | | | | | | | | | | | | | |


Clinical Study Protocol: BOS161721-02

 Table 2.
 Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screen <sup>a</sup> | Enroll | | | | Т | reatme | nt Period | d Follow | -iin | | | | Safet | y Follo | w-Un |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | Screen | Emon | | | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | | | 7 | 8 | 9 |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| | | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | -28 to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| General | | | | | | | | | | | | | | | | |
| BOS161721 or placebo dosing | | X | | | X | | X | X | X | X | X | | | | | |
| Injection site reaction assessment <sup>e</sup> | | X | | | X | | X | X | X | X | X | | | X | X | X |
| Targeted physical examination | | | | X | X | X | X | X | X | X | X | | | X | X | X |
| Vital signs (BP, HR, and temperature) <sup>f</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| Urine pregnancy test (women) <sup>g</sup> | | X | | | X | | X | X | X | X | X | | | | | |
| Spot urine for protein/creatinine ratio | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Urinalysis | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Concomitant medication <sup>h</sup> | X | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| AEs and SAEs | | X | | X | X | X | X | X | X | X | X | | | X | X | X |
| BILAG-2004 Index | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLEDAI-2K | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| PGA | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| ACR-28 joint count | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CLASI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| SLICC/ACR<br>Damage Index | | X | | | _ | _ | _ | | | | X | | | | | |


Clinical Study Protocol: BOS161721-02

 Table 2.
 Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screen <sup>a</sup> | Enroll | | | | T | reatme | nt Perio | d Follow | -up | | | | Safet | y Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | | | 7 | 8 | 9 |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| | | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | -28 to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| CCI | | X | | | X | | X | X | X | X | X | | | X | X | X |
| 12-lead ECG <sup>i</sup> | X | X | | | X | | | X | | | | | | | | X |
| Laboratory | | | | | | | | | | | | | | | | |
| CD4+ count | X | X | | X | X | X | | X | | | X | | | | | |
| Clinical laboratory<br>assessments<br>(hematology and | | | | | | | | | | | | | | i | | |
| clinical chemistry) | X <sup>j</sup> | X | | | X | | X | X | X | X | X | | | X <sup>j</sup> | X | X |
| Coomb's test direct <sup>k</sup> | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Total IgG and IgM | X | X | | X | X | X | | X | | | X | | | | | |
| Plasma CCI | X | X | | | X | | X | X | X | X | X | | | X | X | X |
| Plasma CCI & | X | X | | X | X | | X | X | | | X | | | | | |
| Whole blood for leukocyte immunophenotype | X | X | | X | X | | X | X | | | X | | | | | |
| ADA <sup>l</sup> | | X | | X | X | | X | X | | | X | | | | | X |
| nAb <sup>m</sup> | | | | | | | | X | | | X | | | | | |
| pSTAT3 <sup>n</sup> | | X | | | X | X | X | X | | | X | | | | | |
| CCI | | X | | | | | | | | | X | | | | | |
| Whole blood RNA collection | | X | | X | X | | | X | | | | | | | | X |
| CCI | X | X | | | X | | X | X | X | X | X | | | X° | X° | X° |


Clinical Study Protocol: BOS161721-02

Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screen <sup>a</sup> | Enroll | | | | 7 | [reatme | nt Perio | d Follow | -up | | | | Safet | y Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | | 7 | 8 | 9 | | | | | | | |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| | | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | -28 to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | 11 | 12 | 13 |
| CRP | X | | | | | | | X | | | | | | | | X |
| PK Labs <sup>p</sup> | | | | | | | | | | | | | | | | |
| Predose <sup>q</sup> | | X | | | X | | X | X | X | X | X | | | | | |
| Postdose | | | | X | | | | | | | | X | X | X | X | X |

Abbreviations: ACR = American College of Rheumatology; ADA= anti-drug antibody; AE = adverse event; CCl ; BILAG = British Isles Lupus Assessment Group; BP = blood pressure; C = complement; CD4+ = cluster of differentiation 4; CLASI = Cutaneous Lupus Area and Severity Index;

CRP = C-reactive protein; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; CC ; FSH = follicle stimulating hormone; HR = heart rate; HIV = human immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; IL-21 = interleukin 21; IV = intravenous; nAb = neutralizing antibody; PGA = Physician's Global Assessment; PK = pharmacokinetic; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; RNA = ribonucleic acid; RNP = ribonucleoprotein; SAE = serious adverse event; SC = subcutaneous; CC ; SLEDAI-2K = SLE Disease Activity Index 2000; SLICC = Systemic Lupus International Collaborating Clinics; TB = tuberculosis; TDAR = T-cell dependent antigen response.

- Screening assessments will be performed over more than 1 visit.
- If patients have had a TB test and chest x ray within 3 months prior to screening, then these assessments do not need to be repeated during screening. The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 1).
- <sup>c</sup> Cryptosporidium test is required at screening. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- Randomization should occur after patient eligibility has been confirmed. The actual randomization procedure can be completed on Day -1 after eligibility confirmation or the morning of Day 1 prior to dosing for logistical purposes.
- <sup>e</sup> Injection site reaction assessments to be performed predose and at 2 hours postdose.
- f Vital signs will be assessed after the patient has been supine and at rest ≥ 5 minutes. Vital signs will be assessed on Day 1 at predose and at 1 and 2 hours postdose as well as on each of the scheduled outpatient days in the table above. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.
- <sup>g</sup> Urine pregnancy test will be collected on WOCBP prior to study drug administration on dosing visits.
- Concomitant use of oral corticosteroids: A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 1 (randomization day). See Section 5.6.1 for further details.
- ECGs will be performed after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK


Clinical Study Protocol: BOS161721-02

Table 2. Schedule of Assessments - Phase 2 Proof of Concept (POC) Study

| | Screen <sup>a</sup> | Enroll | | | | 1 | reatme | nt Perio | d Follow | -up | | | | Safet | y Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Months | | | | | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | | | 7 | 8 | 9 |
| Weeks | | | 1 | 2 | 4 | 6 | 8 | 12 | 16 | 20 | 24 | 25 | 26 | 28 | 32 | 36 |
| | | | 7 | 15 | 30 | 44 | 60 | 90 | 120 | 150 | 180 | 187 | 195 | 210 | 240 | 270 |
| Days | -28 to -1 | 1 | (± 1) | (± 3) | (± 3) | (± 3) | (± 3) | $(\pm 3)$ | (± 3) | (± 3) | $(\pm 3)$ | $(\pm 3)$ | (± 3) | (± 3) | (± 3) | (± 3) |
| Visit Number | 1 | 2 | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | _ | | 11 | 12 | 13 |

blood draws (Section 7.5).


Clinical laboratory assessments will include a fasting glucose and lipid panel during screening and Week 28

When clinically indicated.

Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.

m nAb is assessed if patient is positive for ADA.

<sup>&</sup>lt;sup>n</sup> Predose (trough) samples only.

Only CCl collected during safety follow-up visits.

PK samples will only be collected at the investigational sites that will be participating in the PK portion of the study.

<sup>&</sup>lt;sup>q</sup> Predose samples occur on study drug administration visit days.

## 5 POPULATION

# 5.1 Participant Recruitment

Advertisements approved by the IRB, and investigator databases, may be used as recruitment procedures for adult men and women with moderately to severely active SLE.

## **5.2** Number of Patients

Approximately 186 male and female patients are planned for enrollment, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Approximately 30 patients will be randomized for the MAD Phase 1b study, and approximately 156 patients will be randomized in the POC Phase 2 study. Note that approximately 30 dropouts are assumed.

# **5.3** Patient Screening

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular individual. Patient eligibility will be reviewed and confirmed by the medical monitor or designee prior to randomization. Screening assessments (see the Schedule of Assessments [Section 4.3]) for this study must be performed between Day -28 and Day -1.

#### 5.4 Inclusion Criteria

Patients who meet the following criteria will be considered eligible to participate in this clinical study:

- 1. Men and women, ages 18 to 70 years, inclusive;
- 2. Patients must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
- 3. Patients must have SLE as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion or Lupus nephritis as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies), either sequentially or simultaneously.
- 4. At screening, patients must have at least 1 of the following:
  - a. Elevated antinuclear antibodies (ANA) ≥ 1:80 via immunofluorescent assay at the central laboratory;
  - b. Positive anti-dsDNA or anti-Smith (Sm) above the normal level as determined by the central laboratory;
  - c. C3 or C4 below normal as determined by central lab.

- 5. At screening, the SLE Disease Activity Index 2000 (SLEDAI-2K) must be ≥ 6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis
    - i. Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia)
    - ii. Points from lupus headache and organic brain syndrome will also be excluded.
- 6. On Day 1, the SLEDAI-2K must be  $\geq$  6, including points from at least 1 of the following clinical components:
  - a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis.
    - i. Excluding parameters which require central laboratory results: (hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia);
    - ii. Points from lupus headache and organic brain syndrome are also excluded.
- 7. Patients must have at least 1 of the following manifestations of SLE, as defined by the BILAG criteria as modified for use in this study, which must be confirmed by the central data reviewer:
  - a. BILAG A or B score in the mucocutaneous body system;
  - b. BILAG A or B score in the musculoskeletal body system due to active polyarthritis defined as follows:
    - i. "BILAG A:" Severe Arthritis, (BILAG item number 41), manifested by observed active synovitis in ≥ 2 joints with marked loss of functional range of movements and significant impairment of basic activities of daily living that has been present on several days cumulatively over the past 4 weeks, including at the time of the screening visit. See APPENDIX 5 for additional detailed specifications.
      - Basic ADLs are defined as the following activities which require assistance or assistive devices, (at least 1 must be present and documented in source):
        - o Ambulation, toileting, grooming- including bathing and dressing; feeding oneself, (and not responsive to steroids up to 10 mg/day, antimalarials, NSAIDs).
    - ii. "BILAG B:" Moderate Arthritis, Tendonitis or Tenosynovitis, (BILAG item number 42), defined as tendonitis/tenosynovitis, or active synovitis in ≥ 1 joint, (observed or throughout history), with some loss of functional range of movements which lead to some loss of functional range of motion as manifested by effects on instrumental ADLs such as:

- Cooking, driving, using the telephone or computer, shopping, cleaning, etc, and has been present on several days over the last 4 weeks, and is present at the time of the screening visit.
- c. If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in the other body systems for a total of 2 "B" BILAG body system scores.
- 8. Patients must be currently receiving at least 1 of the following:
  - a. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to signing consent) of the following permitted steroid-sparing agents:
    - i. Azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate (MTX).
  - b. Prednisone (or prednisone-equivalent) cannot exceed 30 mg/day at screening for a patient to be eligible and must be stable at a maximum of 10 mg/day for at least 5 days prior to Day 1 (randomization) (see APPENDIX 3).
- 9. Women of childbearing potential (WOCBP; see Section 5.7 for full information regarding WOCBP, definition of menopause, and contraception):
  - a. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose;
  - b. Must not be breastfeeding;
  - c. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion;
- 10. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion.
- 11. Patients must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures.

#### 5.5 Exclusion Criteria

Patients presenting with any of the following will not be included in this study:

- 1. Drug-induced SLE, rather than "idiopathic" SLE;
- 2. Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic scleroderma, or vasculitis not related to SLE);
  - a. RA-Lupus overlap (Rupus), and secondary Sjögren syndrome are allowed.
- 3. Any major surgery within 6 weeks of study drug administration, (Day 1), or any elective surgery planned during the course of the study;
- 4. Any history or risk for tuberculosis (TB), specifically those with:
  - a. Current clinical, radiographic, or laboratory evidence of active TB;
  - b. History of active TB;
  - c. Latent TB defined as positive QuantiFERON-TB Gold In-Tube (QFT-G) or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the patient has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the patient has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 1 and continues to receive the prophylactic treatment during study until the treatment course is completed.
- 5. Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed;
- 6. Severe proliferative lupus nephritis, (WHO Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CS;
- 7. Concomitant illness that, in the opinion of the investigator, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary;
  - a. However, treatment for asthma with inhalational CS therapy is allowed.
- 8. Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study. (See Section 5.6 for prohibited concomitant medication);
- 9. Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic antibiotics or hospitalization;
- 10. A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years;
- 11. Chronic viral hepatitis including hepatitis B (HBV) and hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness;
- 12. Cryptosporidium in the stool sample at screening;
- 13. White blood cells (WBC)  $< 1,200/\text{mm}^3 (1.2 \times 10^9/\text{L})$  at screening;
- 14. Absolute neutrophil count (ANC) < 500/mm<sup>3</sup> at screening;
- 15. CD4+ count  $< 500/\mu L$  at screening;
- 16. Platelets < 50,000/mm $^3$  (50  $\times$  10 $^9$ /L) or < 35,000/ mm $^3$  (35  $\times$  10 $^9$ /L) if related to SLE, at screening;
- 17. Hemoglobin < 8 g/dL or < 7 g/dL at screening if due to anemia related to SLE;
- 18. Proteinuria > 3.0 g/day (3000 mg/day) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 mg/mmol);

- 19. Serum creatinine > 2.0 mg/dL at screening or creatinine clearance (CrCL) < 40 ml/minute based on Cockcroft-Gault calculation<sup>39</sup>:
  - GFR = ([1 for male] or [0.85 for female])  $\times$  (140 Age)  $\times$  BW / (72  $\times$  Creatinine)
- 20. Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) > 2 × ULN at screening, unless explicitly related to lupus based on the investigator's judgment;
- 21. Creatinine kinase (CK)  $> 3.0 \times$  ULN at screening, unless it is related to lupus myositis
- 22. Direct bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome);
- 23. Any other laboratory test results that, in the opinion of the Investigator, might place a patient at unacceptable risk for participating in this study;
- 24. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (eg, IgG protein) or molecules made of components of monoclonal antibodies;
- 25. History substance and/or alcohol abuse or dependence within the past 1 year, at the investigator's judgement;
- 26. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision);
- 27. Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
- 28. Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the sponsor or directly involved in the conduct of the trial;
- 29. Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer;
- 30. Recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4 or 5 on the Columbia Suicide severity Rating Scale (C-SSRS);
- 31. Current or pending incarceration;
- 32. Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness.

#### **5.6** Concomitant Medications

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Patients should stay on stable regimen of other

BOS161721 Clinical Study Protocol: BOS161721-02

concomitant medications for the treatment of SLE (eg, analgesics, NSAIDs, statins, ACE inhibitors/ARBs and other antihypertensive drugs), unless changes in these treatments are clinically indicated. Use of any other drugs for non-SLE conditions, including over-the-counter medications and herbal preparations, should remain stable unless change or addition is clinically necessary. Discussion with the medical monitor prior to initiation of new medication is strongly recommended. Any concomitant therapies must be recorded on the eCRF. Prior and concomitant medication use will be recorded for the 30 days prior to screening until the last follow-up visit. In addition, historical treatment for SLE (including immunosuppressant, anti-malarial, corticosteroid, and/or biologic agent) will be recorded for the 48 weeks prior to screening in the eCRF.

#### 5.6.1 Oral Corticosteroid Dose

Prior to randomization, oral CSs (prednisone or prednisone equivalent), may be used in accordance with the investigator's clinical judgment and best standard of care. See APPENDIX 3 for examples of equivalents.

A maximum daily dose of 30 mg/day of oral CS will be acceptable for eligibility for the study, however, the daily dose must be tapered down to a maximum of 10 mg/day for at least 5 days prior to Day 1 (randomization day).

After Day 1 (after initiation of study therapy), no up-titration above 10 mg/day is allowed except for up to 1 CS burst for increased disease activity.

Tapering of steroids during the course of the study will be encouraged and should be evaluated at all visits.

- Once a patient has received the first dose of study drug, prednisone (or prednisone equivalent) may be tapered down at the discretion of the investigator;
  - O Tapering is allowed after randomization except within 8 weeks of the primary (Week 28) and secondary (Week 16) endpoint assessments. Between Week 8 and Week 16, and between Week 20 and Week 28, oral corticosteroid (OCS) doses must be held constant otherwise the patient will be declared a non-responder in efficacy assessments.

A maximum of 1 oral CS "burst" for increased SLE disease activity will be allowed during the study either between Weeks 1 and 8 or between Weeks 16 and 20, according to the following:

- An oral CS "burst" between Week 1 and Week 8; (an increase of ≤ 40 mg/day of prednisone or equivalent), which must be tapered down to a maximum of 10 mg/day within 2 weeks of initiation of the "burst."
  - O Alternatively, a single intramuscular (IM) dose of methylprednisolone (40 mg or equivalent) is permitted;
  - o The course of the oral CS "burst" is not permitted to extend beyond Week 8.

- An oral CS "burst" between Week 16 and Week 20 (an increase of ≤ 20 mg/day prednisone or equivalent), which must be tapered down to a maximum of 10 mg/day within 2 weeks of initiation of the "burst".
  - o Alternatively, a single IM dose of methylprednisolone (40 mg or equivalent) is permitted.

Treatment with inhalational CS therapy (eg, for asthma), or by any other route, is allowed. Other concomitant medications for SLE need to be taken at stable doses as per the inclusion criteria (Section 5.4).

#### **5.6.2** Other Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken prior to study drug administration in the study are described below, and washout requirements are provided in APPENDIX 4. Medications taken within 30 days prior to screening must be recorded on the eCRF.

- 1. Prior exposure to BOS161721;
- 2. Patients who have received treatment with anti-CD20 monoclonal antibodies within 6 months of screening; recovery of B cells (CD19+) must be documented (record absolute number of CD19+ B cells);
- 3. Patients who have received treatment with cyclophosphamide within the 1 year prior to screening;
- 4. Patients who have received treatment with cyclosporine (with exception of ophthalmic use), any other calcineurin inhibitor or other immunosuppressive medication not specified in the inclusion criteria (oral or topical) within 3 months of screening;
- 5. Patients who are currently receiving or are scheduled to receive plasmapheresis or lymphapheresis therapy, or have received such therapy within 8 weeks prior to screening;
- 6. Patients who have received any live vaccines within 30 days of screening. Note: Furthermore, live vaccines should not be used during the course of the study and within the 2 months following last dose. Other inactivated vaccines such as tetanus, etc, may be used according to local guidelines during treatment period;
- 7. Patients who are scheduled or anticipated to have elective surgery during the course of the study;
- 8. Initiation of new immunosuppressant or anti-malarial agent is not permitted. Note: Dose reduction or replacement may be allowed due to intolerability or shortage for patients on a stable dose prior to study initiation.

# **5.7** Women of Childbearing Potential

WOCBP is defined as any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) and is not postmenopausal.

See Section 5.7.2 for detailed information regarding contraceptive requirements for WOCBP.

# **5.7.1** Determination of Menopause

Menopause is defined as at least 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes. Women under the age of 55 years must have a documented serum FSH level > 40 mIU/mL at screening to confirm menopause.

## 5.7.2 Contraception

WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 30 days (duration of ovulatory cycle) for a total of 36 weeks after treatment completion.

Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug BOS161721 plus 90 days (duration of sperm turnover) for a total of 44 weeks after treatment completion.

Investigators shall counsel WOCBP and men who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and men who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, patients must agree to the use of 1 method of highly effective contraception from the following:

- Male condoms with spermicide;
- Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by patients who are WOCBP or a male patient's WOCBP partner. Women who are partner of men who are patients participating in the study may use hormone-based contraceptives as 1 of the acceptable methods of contraception since they will not be receiving study drug.
- IUDs, such as ParaGard®;
- Vasectomy;
- Complete abstinence, defined as complete avoidance of heterosexual intercourse, is an
  acceptable form of contraception. Women who are abstinent while participating in the study
  must continue to have pregnancy tests. Acceptable alternate methods of highly effective
  contraception must be discussed in the event that the patient chooses to forego complete
  abstinence.

Azoospermic men and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing.

#### 5.8 Deviation from Inclusion/Exclusion Criteria

Deviation from the inclusion or exclusion criteria will not be allowed. If deviation of inclusion/exclusion criteria is discovered after randomization, the investigator should contact the medical monitor for discussion. A decision will be made whether to allow a patient continue or withdrawal from the study medication.

See Section 7.8 for additional details.

### 5.8.1 Patient Withdrawal and Replacement

See Section 6.5 for reasons for removal from the trial. Withdrawn patients may be replaced during the MAD study after discussion between the principal investigator or designee and sponsor.

### **5.8.2** Exception for Non-Responders

Patients will be classified as non-responders if they (1) receive a second rescue medication at any time in the study or (2) take rescue medications between Week 8 and Week 16 or between Week 20 and Week 28 (as described in Section 5.6.1). If a patient has been deemed a non-responder, they will discontinue from treatment and all End of Treatment assessments will be performed. The patient will then enter the safety follow-up period. The use of rescue medications in the case of non-responders is not to be considered a protocol violation (exclusion criteria 8). Protocol violations will be identified based on blinded data prior to unblinding the final analysis dataset.

BOS161721 Clinical Study Protocol: BOS161721-02

### 6 STUDY PROCEDURES

Refer to the eCRF completion guidelines for data collection requirements and documentation of study assessments/procedures.

# 6.1 Screening

Screening will be the same for both the MAD and POC studies. Screening for the POC study cannot begin until the POC dose decision has been made.

Screening will take place from Day -28 to Day -1, and assessments may be performed over more than 1 visit. Confirmation that the most current IRB/IEC approved informed consent form (ICF) has been signed must occur before any study-specific screening procedures are performed. Procedures that are part of standard of care are not considered study-specific procedures and may be performed prior to informed consent and used to determine eligibility.

All screened patients will be assigned a unique screening number. The screening number will include a 3-digit site number and a 4-digit sequential number to identify patients from the time of screening. Only eligible patients who are confirmed by central review as meeting the inclusion/exclusion criteria listed in Section 5.4 and Section 5.5 will be enrolled in the study. Screened patients who drop out of the clinical study before randomization will be recorded as screen failures. If rescreening occurs, the site will assign a new screening number.

Specific procedures at the screening visit will include:

- Medical history documentation;
- Review of inclusion and exclusion criteria;
  - o Patient medical records must contain documentation of SLE diagnosis;
  - o C-SSRS.
- Concomitant medication documentation;
- Demographics;
- Full physical examination;
- Vital signs;
- Laboratory evaluations:
  - o Hematology and clinical chemistry;
  - Serology (Hepatitis B and C; HIV-1/2 combination);
  - o TB test

- o CRP
- o Direct Coomb's test (if indicated)
- CD4+ count, total IgG and IgM levels, plasma CO , plasma CO , whole blood for leukocyte immunophenotype; CO ;
- Serum pregnancy test (WOCBP);
- o FSH and estradiol (postmenopausal women)
- Spot urine for protein/creatinine ratio;
- o Urinalysis.
- Stool sample
- 12-lead ECG;
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, Physician's Global Assessment (PGA) of disease activity.

Screening procedures are listed in the Schedule of Assessments (Section 4.3), and details are provided in Section 7.

## **6.1.1** Retesting During Screening Period

A single retesting of laboratory parameters and/or other assessments during the screening period is permitted (in addition to any parameters that require a confirmatory value) only if:

- medically indicated;
- there is evidence a laboratory sample was mislabeled, inadequately processed, and/or deteriorated in transit to the central laboratory.

Any new result will override the previous result (ie, the most current result prior to randomization) and is the value by which study inclusion/exclusion will be assessed, as it represents the patient's most current clinical state. This will also apply to patients who are being rescreened.

# 6.2 Enrollment/Randomization and Day 1 Treatment

Randomization should occur after patient eligibility for enrollment has been confirmed by the central eligibility review.

The study site will obtain a randomization number when registering the patient in IWRS. All patients will receive BOS161721 or placebo according to the kit number assigned by the IWRS randomization scheme.

After randomization, procedures include:

- PROs: CCl ;
- C-SSRS;
- Laboratory evaluations:
  - Hematology and clinical chemistry
  - Direct Coomb's test (if indicated)
  - o CD4+ count, total IgG and IgM levels, plasma CCl , plasma CCl , whole blood for leukocyte immunophenotype;
  - o ADA;
  - o pSTAT3 (predose [trough] samples only in Phase 2);
  - o CCI ;
  - Whole blood RNA collection;
  - o <mark>CCI</mark>;
  - o See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies;
  - o Urine pregnancy test will be collected on WOCBP prior to study drug administration;
  - Spot urine for protein/creatinine ratio;
  - Urinalysis.
- Concomitant medication documentation;
- Documentation of AEs and SAEs (see Section 7.2.2.5 on SAE reporting requirements);
- Full physical examination;
- Vital signs (prior to PK blood draw, predose, and at 1 and 2 hours postdose on Day 1);
- 12-lead ECG (prior to PK blood draw);
- SLE-related indices (BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, PGA);
- SLICC/ACR damage index;
- Study drug administration;

- o Administration of BOS161721 or placebo will take place on-site, and is discussed in Section 8.3.
- Injection site reaction assessment, predose and 2 hours postdose.

Procedures on Day 1 are listed in the Schedule of Assessments (Section 4.3), and details are provided in Section 7.

All patients who are enrolled, randomized, and receive study drug, or undergo study-specific procedures should reconsent with any updated versions of IRB/IEC approved informed consents during study participation as applicable and per institutional guidelines.

## 6.3 Treatment Period/Follow-Up Visits

See Section 4.3 for allowable windows for each visit. The following procedures will be performed at every study drug administration visit (Weeks 4, 8, 12, 16, 20, and 24) and follow-up visits during the treatment period (Weeks 2 and 6):

- Targeted physical examination;
- Vital signs (prior to PK blood draw);
- Concomitant medication documentation;
- Documentation of AEs and SAEs (see Section 7.2.2.5 on SAE reporting requirements).

The following assessments will be performed only at Weeks 4, 8, 12, 16, 20, and 24:

- PROs: CCl ;
- Urine pregnancy tests will be collected on WOCBP prior to study drug administration;
- Injection site reaction assessments will be performed predose and 2 hours postdose;
- Direct Coomb's test (if indicated);
- Spot urine for protein to creatinine ratio;
- Urinalysis;
- CCI
- Plasma CC ;
- PGA, BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, and the CLASI will be completed.
- In addition the following assessments will be completed:

- SLICC/ACR Damage Index will be completed at Week 24 (Visit 10).
- C-SSRS will be completed at Weeks 12 and 24 (Visits 7 and 10);
- ECGs will be performed at Weeks 4 and 12 (Visits 4 and 7) prior to PK blood draw.
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies, respectively.
- Hematology and chemistry assessments will be performed at Weeks 4 and 6 (Visits 4 and 5) for the MAD study, only, and at Weeks 8, 12, 16, 20, and 24 (Visits 6 through 10) for both studies.
- The CD4+ count and total IgG and IgM levels will be assessed at Weeks 2, 4, 6, 12, and 24 (Visits 3, 4, 5, 7, and 10).
- Plasma **CCl** & **CCl** and ADA, and whole blood for leukocyte immunophenotype will be assessed at Weeks 2, 4, 8, 12, and 24 (Visits 3, 4, 6, 7, and 10).
- pSTAT3 will be assessed at Weeks 4, 6, 8, 12, and 24 (Visits 4, 5, 6, 7, and 10).
- Whole blood RNA will be collected at Weeks 2, 4, and 12 (Visits 3, 4, and 7).
- CRP will be measured at Week 12 (Visit 7), and nAb will be assessed if patient is positive for ADA at Weeks 12 and 24 (Visits 7 and 10).
- CCl will be assessed at Week 24 (Visit 10).

# 6.4 Safety Follow-Up Visits

Safety follow-up visits will take place at Weeks 28, 32, and 36 (Visits 11, 12, and 13). These visits will include the following:

- PROs: CCI ;
- Documentation of AEs and SAEs (see Section 7.2.2.5 on SAE reporting requirements);
- Injection site reactions;
- Targeted physical examination;
- Vital signs (prior to PK blood draw);
- Spot urine for protein/creatinine ratio and urinalysis;
- Concomitant medication documentation;
- BILAG-2004 Index, SLEDAI-2K, ACR-28 joint count, CLASI, and PGA;

- Clinical laboratory assessments (hematology and clinical chemistry);
- Direct Coomb's test (if indicated);
- Plasma CCI ;
- CCI
- pSTAT3 (Week 36 only for MAD study);
- 12-lead ECG (Week 36 only, prior to PK blood draw);
- CRP (Week 36 only);
- ADA (Week 36 only);
- Whole blood RNA collection (Week 36 only);
- See Table 1 and Table 2 for details of PK sampling in the MAD and POC studies, respectively.

#### 6.5 Premature Discontinuation

While patients are encouraged to complete all study evaluations, they may withdraw from the study at any time and for any reason. Every effort will be made to determine why any patient withdraws from the study prematurely. If the patient is unreachable by telephone, a registered letter, at the minimum, should be sent to the patient requesting him/her to contact the clinic.

All patients who withdraw from the study with an ongoing AE or SAE must be followed until the end of study or until the event is resolved or deemed stable, respectively.

If a patient withdraws prematurely after dosing, an end of treatment (EOT) visit should be performed (Visit 10) and a last follow-up visit 90 days after dosing should be scheduled (Visit 13). Safety follow-up visit procedures based on the Schedule of Assessments (see Section 6.4).

Patient participation may be terminated prior to completing the study and the reason recorded as follows:

- AE/SAE;
- Protocol deviation;
- Lost to follow-up;
- Patient withdraws consent at their own request;
- Investigator decision;

• Decision by sponsor (other than AE/SAE, protocol deviation, or lost to follow-up).

Withdrawn patients may be replaced after discussion between the investigator or designee and sponsor.

#### 7 ASSESSMENTS

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances, outside of the control of the investigator, which may make it unfeasible to perform the test. In these cases, the investigator will take all steps necessary to ensure the safety and wellbeing of the patient. When a protocol required test cannot be performed the investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. All protocol violations are entered directly into the eCRFs.

# 7.1 Medical History, Demographic and Other Baseline Information

The medical history comprises:

- General medical history;
- Documentation of SLE diagnosis;
- Historical medication therapy for SLE.

The following demographic information will be recorded:

- Age;
- Ethnic origin (Hispanic/Latino or not Hispanic/not Latino);
- Race (White, American Indian/Alaska Native, Asian, Native Hawaiian or other Pacific Islander, Black/African American);
- Height (without shoes, in cm);
- Body weight, without shoes (kg);
- Body mass index (BMI [kg/m²]).

Other baseline characteristics will be recorded as follows:

- Concomitant medication documentation (see Section 5.6);
- Status of child bearing potential and contraception.

## **7.2** Safety Assessments

## 7.2.1 Laboratory Assessments

Laboratory tests will be performed at times defined in the Schedule of Assessments (Section 4.3). Patient eligibility will be determined based on these tests at screening. Unscheduled clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

A central laboratory will be used (with the exception of urine pregnancy tests and stool analysis) to ensure accuracy and consistency in test results. The central laboratory will transmit all results for protocol tests, scheduled and unscheduled, to the clinical data base. Laboratory/analyte results that could unblind the study (ie, biomarker results) will not be reported to investigative sites or other blinded personnel until the study has been unblinded. Urinalysis will be performed on midstream, clean catch specimens. Some biomarkers listed above will not be drawn at some sites due to geographical logistical challenges. See the laboratory manual for details.

Table 3. Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other Safety Tests |
|---|---|---|---|
| Hemoglobin | BUN | рН | Spot urine for protein/creatinine ratio |
| Hematocrit | Creatinine | Glucose (qual) | FSH <sup>b</sup> |
| RBC count | Glucose (fasting) | Protein (qual) | Estradiol <sup>b</sup> |
| RDW | Calcium | Blood (qual) | Urine pregnancy test <sup>c</sup> |
| MCV | Sodium | Ketones<br>Nitrites | QuantiFERON®-TB Gold In-Tube test<br>(QFT-G) |
| MCH | Potassium | | |
| MCHC | Chloride | Leukocyte esterase | Serology <sup>d</sup> (Hepatitis B and C; HIV-1/2 |
| Platelet count | Total CO <sub>2</sub> (bicarbonate) | Urobilinogen | combination) |
| WBC count | AST, ALT | Urine bilirubin | Stool sample <sup>e</sup> |
| CD4+ count | Total bilirubin | Microscopy <sup>a</sup> | |
| Total neutrophils (Abs) | Alkaline phosphatase | 17 | |
| Eosinophils (Abs) | Creatine kinase | | |
| Monocytes (Abs) | Uric acid | | |
| Basophils (Abs) | Albumin | | |
| Lymphocytes (Abs) | Total cholesterol | | |
| Reticulocytes (%) | (fasting) | | |
| , , | LDL-C (fasting) | | |
| | HDL-C (fasting) | | |
| | Triglycerides (fasting) | | |
| | Total protein | | |
| PT/IN Addi | PT/INR | | |
| | Additional Tests <sup>f</sup><br>(potential Hy's Law) | | Immunogenicity, PD and other<br>Biomarker Tests |
| | AST, ALT (repeat) | | ADA |
| | Total bilirubin (repeat) | | $nAb^g$ |
| | Albumin (repeat) | | pSTAT3 (predose [trough] samples |
| | Alkaline phosphatase | | only, in Phase 2) |
| | (repeat) | | Total IgG & IgM |
| | Direct bilirubin | | Plasma <mark>CC</mark> |
| | Indirect bilirubin | | Plasma CCI & CCI |
| | GGT | | Whole blood for leukocyte |
| | | | immunophenotype and RNA |
| | | | CCI |
| | | | Antibodies CCI |
| | | | CRP |
| | | | Direct Coomb's test <sup>h</sup> |

Abbreviations: Abs = absolute; ADA = anti-drug antibody; ALT = alanine aminotransferase;

; CCl ; AST = aspartate aminotransferase; BUN = blood urea nitrogen; C = complement; CD4+ = cluster of differentiation 4; CRP = C-reactive protein;

dsDNA = double-stranded deoxyribonucleic acid;; FSH = follicle stimulating hormone; GGT = gamma-glutamyltransferase; HDL-C = high-density lipoprotein cholesterol; HIV = human

immunodeficiency virus; IgG = immunoglobulin G; IgM = immunoglobulin M; INR = international normalized ration; IL-21 = interleukin 21; LDL-C = low-density lipoprotein cholesterol; MCH = mean corpuscular hemoglobin;

MCHC = mean corpuscular hemoglobin concentration; MCV = Mean corpuscular volume; nAb = neutralizing antibody; pSTAT3 = phosphorylated signal transducer and activator of transcription 3; PT = prothrombin time; qual = qualitative; RBC = red blood cell; RDW = RBC distribution width; RNA = ribonucleic acid;

RNP = ribonucleoprotein; SAE = serious adverse event; SC = subcutaneous; CC

; TB = tuberculosis.

BOS161721 Clinical Study Protocol: BOS161721-02

Table 3.Laboratory Tests

| Hematology Chemistry Urinalysis Other Safety | Tests |
|----------------------------------------------|-------|

- a. On all urine samples.
- b. At screening only, in women who are amenorrheic for at least 12 consecutive months and under 55 years old.
- c. For WOCBP.
- d. Screening only.
- At screening, and if a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.
- Additional testing for potential Hy's Law cases only (See Section 7.2.2.6.3).
- g. If patient is positive for ADA.
- h. If clinically indicated.

# 7.2.1.1 Pregnancy testing

For WOCBP, a serum pregnancy test will be performed at screening. Following a negative serum pregnancy result at screening, appropriate contraception must be commenced or continued and a further negative urine pregnancy test results will then be required at the baseline visit before the patient may receive the investigational product. Urine pregnancy tests will also be routinely repeated at study drug administration visits (Visits 2, 4, 6, 7, 8, 9, and 10) prior to study drug administration, and additionally whenever 1 menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive pregnancy test or confirmed pregnancy, the patient will be withdrawn from study drug but may remain in the study for safety monitoring.

See Section 7.2.2.7.1 for information on reporting of pregnancies as AEs/SAEs during the study.

### 7.2.1.2 Tuberculosis Screening

During the screening period, it must be determined and documented that a patient does not have evidence of active or latent or inadequately treated TB per the exclusion criteria (Section 5.5). The results of TB screening, which includes the QuantiFERON®-TB Gold In-Tube (QFT-G) test and a chest x-ray, conducted in the 3 months prior to screening or during the screening period must be documented in study records prior to randomization (Day 1).

# 7.2.1.2.1 Mycobacterium Tuberculosis Testing Using QuantiFERON Test<sup>40</sup>

QuantiFERON®-TB Gold In-Tube (QFT-G) is an in vitro diagnostic test using a peptide cocktail simulating ESAT-6, CFP-10, and TB 7.7 proteins to stimulate cells in heparinized whole blood. Detection of INFγ performed by enzyme-linked immunosorbent assay (ELISA) is used to identify in vitro responses to these peptide antigens that are associated with Mycobacterium tuberculosis infection. QFT-G is an indirect test for M. tuberculosis infection (including disease) and is intended for use in conjunction with risk assessment, radiography and other medical and diagnostic evaluations.

Test results will be reported as positive, negative, or indeterminate. A negative QFT-G test result is required to meet the inclusion criterion. In the case of an indeterminate result, repeat tests should be permitted for the purpose of determining eligibility of patients to enroll in this

study. If a repeat test is indeterminate again, the patient is a screen failure. The procedure for using this test and interpreting the results will be described fully in the laboratory manual, which will be provided to investigators.

#### **7.2.2** Adverse Events

#### 7.2.2.1 Definitions

An AE is defined as any untoward medical occurrence experienced by a study patient, whether or not considered drug related by the principal investigator.

AEs are unfavorable changes in a general condition, subjective or objective signs or symptoms, worsening of pre-existing concomitant disease, and clinically significant abnormality in laboratory parameters observed in a patient in the course of a clinical study.

Non-serious SLE manifestations or abnormal laboratory results related to SLE disease activity would not be recorded as AEs unless they meet the definition for SAEs (Section 7.2.2.5).

## **7.2.2.2** Recording of Adverse Events

AEs should be collected and recorded for each patient from the date of the first dose of study drug until the end of their participation in the study, including the safety follow up period.

AEs may be volunteered spontaneously by the study patient, or discovered by the study staff during physical examinations or by asking an open, nonleading question such as 'How have you been feeling since you were last asked?' All AEs and any required remedial action will be recorded on the Adverse Events eCRF and Safety Adverse Event Form. The details of the AE, date of AE onset (and time, if known), date of AE outcome (and time, if known), and action taken for the AE will be documented together with the principal investigator's assessment of the seriousness of the AE and causal relationship to the study drug and/or the study procedure.

All AEs should be recorded individually, using diagnostic terms where possible. If the diagnosis is not established, individual symptoms may be reported. The AEs will subsequently be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

### 7.2.2.3 Severity of Adverse Events

Each AE will be assessed by the principal investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 criteria. <sup>41</sup> When changes in the severity (grade) of an AE occur more frequently than once a day, the maximum severity for the event should be noted for that day. Any change in severity of signs and symptoms over a number of days will be captured by recording a new AE, with the amended severity grade and the date (and time, if known) of the change.

## 7.2.2.4 Causality of Adverse Events

The principal investigator will assess the causal relationship between BOS161721 or placebo and the AE. One of the following categories (Table 4) should be selected based on medical judgment, considering the definitions below and all contributing factors.

BOS161721 Clinical Study Protocol: BOS161721-02

| Table 4. | Causality Definitions |
|---|---|
| Related | A clinical event, including laboratory test abnormality, occurs in a plausible time relationship to treatment administration and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (dechallenge <sup>a</sup> ) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge <sup>b</sup> procedure if necessary. |
| Unrelated | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative dechallenge and rechallenge information. Typically explained by extraneous factors (eg, concomitant disease, environmental factors, or other drugs or chemicals). |

Dechallenge: Upon discontinuation of a drug suspected of causing an AE, the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation (positive dechallenge), or the symptoms continue despite withdrawal of the drug (negative dechallenge). Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia).

Rechallenge: Upon re-administration of a drug suspected of causing an AE in a specific patient in the past, the AE recurs upon exposure (positive rechallenge), or the AE does not recur (negative rechallenge).

An unexpected adverse drug event is any adverse drug event for which the specificity or severity is not consistent with the current IP.

#### 7.2.2.5 Seriousness of Adverse Events

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death;
- Is life threatening; this means that the patient was at risk of death at the time of the event; it does not mean that the event hypothetically might have caused death if it were more severe;
- Requires hospitalization or prolongation in existing hospitalization;
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions;
- Is a congenital anomaly or birth defect;
- Is another important medical event (see below).

Important medical events that do not result in death, are not life threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such events are:

• Intensive treatment in an emergency room or at home for allergic bronchospasm;

- Blood dyscrasias or convulsions that do not result in inpatient hospitalization;
- Development of drug dependency or drug abuse.

Hospitalization for elective surgery or routine clinical procedures that are not the result of AE (eg, elective surgery for a pre-existing condition that has not worsened) need not be considered SAEs. If anything untoward is reported during the procedure, that occurrence must be reported as an AE, either 'serious' or 'nonserious' according to the usual criteria.

Suspected unexpected serious adverse reactions (SUSARs) are AEs that are associated with the use of the drug and are serious and unexpected.

## **7.2.2.6** Adverse Events of Special Interest

AEs of special interest in this study include the following:

- 1. Anaphylaxis and serious allergic reactions;
- 2. Injection site reaction, including erythema, pain, and induration;
- 3. Drug Induced Liver Injury (DILI) assessed following Hy's Law;
- 4. Malignancy;
- 5. Opportunistic infections such as disseminated histoplasmosis, cryptococcosis, and disseminated tuberculosis;
- 6. Cryptosporidiasis.

#### 7.2.2.6.1 Anaphylaxis and Serious Allergic Reactions

Anaphylaxis will be defined according to the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria. <sup>42</sup> In the event of anaphylactic reaction or severe/serious hypersensitivity/allergic reaction, the patient must discontinue IP and emergency resuscitation measures implemented. In case of other mild to moderate hypersensitivity reaction, depending on the severity, the investigator may manage in accordance with the standard-of-care.

Anaphylaxis is highly likely when any one of the following 3 criteria is fulfilled:

- 1. Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (eg, generalized hives, pruritus, or flushing, swollen lips-tongue-uvula) and at least 1 of the following:
  - a. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow [PEF], hypoxemia)
  - b. Reduced blood pressure or associated symptoms of end-organ dysfunction (eg, hypotonia [collapse], syncope, incontinence)
- 2. Two or more of the following that occur rapidly after exposure to a likely allergen for that patient (minutes to several hours):

- a. Involvement of the skin-mucosal tissue (eg, generalized hives, itch-flush, swollen lips-tongue-uvula)
- b. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)
- c. Reduced blood pressure or associated symptoms (eg, hypotonia [collapse], syncope, incontinence)
- d. Persistent gastrointestinal symptoms (eg, crampy abdominal pain, vomiting)
- 3. Reduced blood pressure after exposure to known allergen for that patient (minutes to several hours):
  - a. Systolic blood pressure of less than 90 mm Hg or greater than 30% decrease from the patient's baseline.

## 7.2.2.6.2 Injection Site Reactions

Injection site reactions are to be captured and reported as AEs. These may include injection site erythema, pain, and induration. The investigator should provide a clear description of the observed or reported AE including location and severity. All concomitant treatments used to treat injection site reactions should be recorded and captured in the eCRF, together with the AE of injection site reactions.

## 7.2.2.6.3 Potential Drug-Induced Liver Injury

Abnormal values in AST and/or ALT levels concurrent with abnormal elevations in total bilirubin level that meet the criteria outlined below in the absence of other causes of liver injury are considered potential cases of DILI, and as potential Hy's Law cases, and should always be considered important medical events. If symptoms compatible with DILI precede knowledge of serum chemical test abnormalities, liver enzyme measurements should be made immediately, regardless of when the next visit or monitoring interval is scheduled. In some cases, symptoms may be an early sign of injury and although typically less sensitive than serum enzyme elevations, they may indicate a need for prompt serum testing. An increase in liver enzymes should be confirmed by a repeated test within 48 to 72 hours following the initial test, prior to reporting of a potential DILI event. Patients will continue to have weekly or biweekly liver enzyme measurements until resolution or levels return to baseline.

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 7.2.2.7.2 for reporting details).

Potential DILI is defined as:

1. ALT or AST elevation  $> 3 \times ULN$ 

AND

2. Total bilirubin > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)

**AND** 

3. No other immediately apparent possible causes of Alt or AST elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic.

The patient should return to the investigational site and be evaluated as soon as possible, include laboratory tests, detailed history, and physical assessment. In addition to repeating measurements of AST and ALT, laboratory tests should include albumin, CK, total bilirubin, direct and indirect bilirubin, GGT, prothrombin time (PT)/International Normalized Ratio (INR), and alkaline phosphatase. A detailed history, including relevant information, such as review of ethanol, acetaminophen, recreational drug and supplement consumption, family history, occupational exposure, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and work exposure, should be collected. Further testing for acute hepatitis A, B, or C infection and liver imaging (eg, biliary tract) may be warranted. All cases confirmed on repeat testing as meeting the laboratory criteria defined above, with no other cause for liver function test (LFT) abnormalities identified at the time should be considered potential Hy's Law cases irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal LFTs. Such potential Hy's Law cases should be reported as SAEs.

Study drug discontinuation is considered if there is marked serum AST or ALT elevation or evidence of functional impairment (as indicated by rising bilirubin or INR, which represent substantial liver injury) that is related to study drug. Discontinuation of treatment should be considered if:

- ALT or AST  $> 8 \times ULN$ ;
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks;

Discontinuation of treatment must occur if:

- ALT or AST >3 × ULN and (total bilirubin > 2 × ULN or INR > 1.5);
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%).

## 7.2.2.6.4 Malignancy

The identification of a malignancy event will be made by the study site and communicated to the sponsor or designee. AEs should be reported as serious per the criteria in Section 7.2.2.5.

After the first dose of study drug, when there is a decision to biopsy a potentially malignant tumor, lymph node, or other tissue, the investigator and/or consultant(s) should contact the sponsor clinicians or designee to discuss the issue and any decisions as soon as possible.

## 7.2.2.6.5 Specific Infections

Any diagnosis or suggested diagnosis of opportunistic infections such as disseminated histoplasmosis, cryptococcosis, shingles, disseminated herpes simplex, or disseminated tuberculosis will be recorded as AEs of special interest.

Cryptosporidiosis is also considered an AE of special interest. Patients will be evaluated for cryptosporidium in the stool at screening, and as clinically indicated (eg, watery diarrhea) during the study. If a patient develops diarrhea during the study a stool sample must be provided to test for ova, parasites, and cryptosporidium.

## 7.2.2.7 Reporting of Adverse Events

AE reporting will be carried out in accordance with applicable local regulations, including regulatory agency and IRB reporting requirements.

Each AE is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 7.2.2.7.2.

## 7.2.2.7.1 Reporting of Pregnancy

As information is available, a pregnancy diagnosed during the study will be reported within 24 hours to the sponsor via the Pregnancy Notification and Outcome Form, including pregnancy in female patients who received study drug and female partners of male study patients who received study drug. The pregnancy should be followed to term and/or outcome and this outcome should also be reported to the sponsor via the Pregnancy Notification and Outcome Form. Pregnancy itself is not regarded as an AE or SAE unless there is complication.

In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an AE or SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live born, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion;
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as serious adverse events when the investigator assesses the neonatal death as related or possibly related to exposure to investigational product.

# 7.2.2.7.2 Reporting of Serious Adverse Events

The principal investigator is responsible for providing notification to the sponsor of any SAE via the Safety Adverse Event Form, whether deemed study drug related or not, that a patient experiences during their participation in this study within 24 hours of becoming aware of the event.

If an SAE is fatal or life threatening, notification to the sponsor must be made aware immediately, irrespective of the extent of available AE information. This timeframe also applies to additional new information (follow-up) on previously forwarded SAE reports as well as to the initial and follow-up reporting of exposure during pregnancy and exposure via breastfeeding cases. In the rare event that the investigator does not become aware of the occurrence of an SAE immediately (eg, if an outpatient study patient initially seeks treatment elsewhere), the investigator is to report the event within 24 hours after learning of it and document the time of his/her first awareness of the AE.

The principal investigator will review each SAE and evaluate the intensity and the causal relationship of the event to the study drug. All SAEs will be recorded from the time of first dose of study drug through the safety follow-up period (up to Week 36). SAEs occurring after the final follow-up visit and coming to the attention of the principal investigator must be reported only if there is (in the opinion of the principal investigator) reasonable causal relationship with the study drug.

As a minimum requirement, the initial notification should provide the following information:

- Study number;
- Patient number;
- Details of the SAE (verbatim details are sufficient for immediate notification);
- Criterion for classification as 'serious';
- Causality assessment (which may be updated in a follow-up report when sufficient information is available to make this classification).

Initial reports of SAEs must be followed later with detailed descriptions, including clear photocopies of other documents as necessary (eg, hospital reports, consultant reports, autopsy reports, etc), with the study patient's personal identifiers removed. All relevant information obtained by the principal investigator through review of these documents will be recorded and submitted to the sponsor within 24 hours of receipt of the information. If a new Safety Adverse Event Form is submitted, then the principal investigator must sign and date the form. The sponsor may also request additional information on the SAE, or clarification of omitted or discrepant information from the initial notification, which the principal investigator or an authorized delegate should submit to the sponsor within 24 hours of the request as possible.

# 7.2.2.7.3 Reporting of Adverse Events of Special Interest

AEs of special interest will be reported to safety immediately or within 24 hours of the site becomes aware of the event and recorded as such on the Adverse Events eCRF and Safety Adverse Event Form.

Potential DILI will be reported based on specifications mentioned in Section 7.2.2.6.3.

Each AE of special interest is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate, and is further outlined in Section 7.2.2.7.2.

# **7.2.2.8** Follow Up of Adverse Events

All AEs will be followed up through the safety follow-up visits. All SAEs experienced by a patient, irrespective of the suspected causality, will be monitored until the event has resolved, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the principal investigator and medical monitor, until there is a satisfactory explanation for the changes observed, or until the patient is lost to follow-up.

See Section 7.2.2.7.1 for details related to follow-up of pregnancy. See Section 7.2.2.6.3 for details related to follow-up of potential DILI. See Section 7.2.2.6.4 for details related to follow-up of malignancy.

## 7.2.3 Vital Signs

Vital signs (blood pressure, heart rate, and body temperature) will be assessed as specified in the Schedule of Assessments (Section 4.3). Vital signs will be assessed on Day 1 at predose and at 1 and 2 hours postdose, as well as on each of the scheduled visit days during the study. Supine BP and heart rate recordings will be made after the patient has been recumbent and at rest  $\geq 5$  minutes. When the timing of these measurements coincides with a blood collection, vital signs should be obtained prior to the time of the blood collection.

#### 7.2.4 12-Lead Electrocardiograms

ECG will be performed at screening, and Visits 2, 4, and 7, and 13. ECG recording will initiate after the patient has been supine for at least 5 minutes. On days of PK blood draws, the ECG will be collected before scheduled PK blood draws, though timing will be such that PK draws are collected on their scheduled times where possible.

The ECG will include all 12 standard leads and a Lead II rhythm strip on the bottom of the tracing. The ECG will be recorded at a paper speed of 25 mm/second. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QT interval corrected for heart rate using Fridericia's formula (QTcF).

All ECGs must be evaluated by a qualified physician or qualified designee for the presence of abnormalities and will be captured electronically and retained for future evaluation if required, up to the time of the clinical study report (CSR) completion.

## 7.2.5 Physical Examinations

The full physical examination will be completed at screening and Visit 2. It includes an assessment of general appearance and evaluation of head, eyes, ears, nose, mouth, throat, neck, thyroid, lymph nodes, and extremities, and dermatologic, respiratory, cardiovascular, gastrointestinal, musculoskeletal, neurologic, and psychiatric systems.

The targeted (limited) physical examination will be completed at Visits 3 through 13. It includes evaluation of patient complaints and SLE disease-related issues, and will exclude the genitourinary system.

#### 7.2.6 C-SSRS

The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed by Columbia University researchers for the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening. 43

The C-SSRS evaluation will be performed at screening, Visit 2 (Day 1) and at Visits 7 and 10 (Weeks 12 and 24, respectively). Patients with recent (within the past 12 months) or active suicidal ideation or behavior based on patient responding "yes" to question 3, 4, or 5 is exclusionary at screening will be excluded from the study. Patients with recent or active suicidal ideation or behavior at subsequent study visits will have responses to the C-SSRS reviewed in detail to assess patient risk, and appropriate consultative mental health services will be provided.

### 7.2.7 Injection Site Reactions

Patients will be monitored for local injection site reactions at dosing administration visits, Visits 2 (Day 1), Visit 4 (Week 4), and Visits 6 through 10 (Weeks 8, 12, 16, 20, and 24). Patients will also be monitored for local injection site reactions at the safety follow-up visits, Visits 11, 12, and 13 (Weeks 28, 32, and 36, respectively). Local injection site reactions will be assessed predose and at 2 hours postdose. Injection site reactions should be managed according to the standard of care. Injection site reactions are to be reported as AEs of special interest (see Section 7.2.2.7.3).

## 7.2.8 Immunogenicity

The serum samples to measure the presence of ADA will be collected as Visits 2, 3, 4, 6, 7, 10, and 13 (Week 0, 2, 4, 8, 12, 24, and 36, respectively). Blood samples (4 mL) to provide approximately 1.5 mL of plasma for anti BOS161721 antibody analysis will be collected into appropriately labeled tubes containing K<sub>2</sub>EDTA. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Day 90 from all patients. Subsequent ADA samples will be collected from all patients but only assayed if the patient had a positive ADA on Day 90.

After the first dose, if a patient tests positive in the validated confirmatory ADA assay, the sample from this patient will be further analyzed in the neutralizing antibody (nAb) assay.

# 7.3 Efficacy Assessments

#### **7.3.1 SLEDAI-2K**

The SLEDAI-2K is a validated instrument that measures disease activity in SLE patients at the time of the visit and in the previous 30 days. It is a global index and includes 24 clinical and laboratory variables that are weighted by the type of manifestation, but not by severity. The total score falls between 0 and 105, with higher scores representing increased disease activity. The SLEDAI-2K has been shown to be a valid and reliable disease activity measure in multiple patient groups. A SLEDAI -2K of 6 or more generally represents moderately to severely active disease. 44

The SLEDAI-2K is completed at screening, at Visit 2, Visit 4, and Visits 6 through 13.

### 7.3.2 BILAG 2004

The BILAG-2004 index is an organ-specific 97-question assessment based on the principle of the doctor's intent to treat. Only clinical features attributable to SLE disease activity are to be recorded and based on the patient's condition in the last 4 weeks compared with the previous 4 weeks. It will be scored as not present (0), improved (1), the same (2), worse (3), or new (4). Disease activity is graded separately for 9 body systems to 5 different grades (A to E) as follows: A ("Active") is very active disease, B ("Beware") is moderate activity, C ("Contentment") is mild stable disease, D ("Discount") is inactive now but previously active, and E ("Excluded") indicates the organ was never involved. A shift from BILAG-2004 Grade A or B to a lower grade indicates a clinically relevant change in disease activity as the BILAG-2004 grades mirror the decision points for treatment interventions.

Only investigators that complete BILAG-2004 training will be allowed to perform the BILAG-2004 assessments. Preferably, the same investigator should evaluate the patient at each BILAG-2004 assessment from screening to study completion. The investigator must maintain documentation with descriptive details supporting the BILAG-2004 scoring (eg, chart, worksheet, clinic notes, and labs) at each visit.

The BILAG-2004 is completed at screening, Visit 2, 4, and 6 through 13. See APPENDIX 5 for detailed specifications.

### 7.3.3 PGA of Disease Activity

The PGA is used to assess investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients".

The PGA is completed at screening, Visit 2, 4, and Visits 6 through 13. When scoring the PGA, the assessor should always look back at the score from the previous visit.

## 7.3.4 Composite Endpoints: SRI-4, SRI-5, SRI-6, and BICLA Response

### **7.3.4.1 SRI-4 Response**

Patients will be evaluated for SRI-4 scores at Week 28, with evaluation for sustained reduction of oral CS ( $\leq$  10 mg/day and  $\leq$  Day 1 dose) between Week 16 and Week 28.

The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. Response based on the SRI-4 is defined by:

1)  $\geq$  4-point reduction in SLEDAI-2K global score, 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B), and 3) no deterioration from baseline in the PGA by  $\geq$  0.3 points. The SRI-4 response in patients with moderate to severe SLE is associated with broad improvements in clinical and patient-reported outcomes. <sup>45</sup>

Each patient, after providing their 28-week SRI-4 response, will be evaluated as either a responder or non-responder.

## 7.3.4.2 SRI-5 and SRI-6 Response

Like the SRI-4, the SRI-5 and SRI-6 are composite indices of SLE disease improvement that consists of scores derived from the SLEDAI-2K and the BILAG 2004 Index. However, the SRI-5 and SRI-6 are computed with a minimal three-point or five-point improvement in SLEDAI-2K being required, respectively. 46

The SRI-5 and SRI-6 are evaluated for response at Week 24, along with a sustained reduction of oral CS ( $\leq$  10 mg/day and  $\leq$  Day 1 dose) between Week 16 and Week 28.

### 7.3.4.3 BICLA Response

The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and PGA. BICLA response is defined as 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (eg, all B [moderate disease] scores falling to C [mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4)  $\leq$  10% deterioration in PGA score and 5) no treatment failure. 44 It is driven primarily by the BILAG, and has been used in Phase 2 and 3 mAb studies. 47

For the endpoints of BICLA response at Week 28, Week 32, and Week 36, patient scores will be completed and response determined.

#### 7.3.5 CLASI Response

The CLASI is a comprehensive tool for assessment of disease activity and damage in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity. <sup>48</sup> Response is defined as 50% improvement from baseline in "A" or "B" scores. This assessment will be applied to all patients as all are required to have cutaneous disease activity.

For the secondary efficacy endpoint of CLASI response at Week 28, patient scores on MAD and POC studies will be compared with baseline for 50% improvement.

#### 7.3.6 ACR-28 Joint Count

The ACR-28 joint count will evaluate the number of tender and swollen joints in the shoulder, elbow, wrist, hand, knee joints. Joints of the feet are excluded. The ACR-28 joint count will be performed at screening, Visit 2, 4, and 6 through 13.

# 7.3.7 Laboratory Assessments

Patients will be evaluated for laboratory parameters as specified in the Schedule of Assessments (Section 4.3), including: Fasting glucose and lipid panels, pSTAT3 (predose samples in Phase 2), total IgG & IgM, complement: CCI, Plasma CCI, whole blood for leukocyte immunophenotype and RNA, CCI, and antibodies: (CCI).

Endpoint analyses will be based on changes from baseline assessments at Week 16 and Week 28.

#### 7.4 Other Variables

## 7.4.1 SLICC/ACR Damage Index

The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in patients with SLE regardless of cause, with demonstrated content, face, criterion, and discriminant validity. It will be performed on Day 1 (Visit 2), and Day 180 (Visit 10).

#### 7.4.2 **PROs**

Patients should be encouraged to complete the PROs at the clinic at the beginning of the study visit prior to any clinical assessments. A member of the staff should be available if a patient requires further instruction and to review the PRO questionnaires for completeness prior to leaving the clinic. The PROs include the CCI and the CCI.



### 7.5 Pharmacokinetic Assessments

During the MAD Phase 1b (all sites) and POC Phase 2 (select sites only) studies, blood samples for PK analysis of BOS161721 or placebo concentration will be collected according to Table 1 and Table 2.

PK parameters include the following:

•  $C_{max}$ ,  $T_{max}$ , AUC,  $t_{\frac{1}{2}}$ , CL,  $V_d$ .

In addition to samples collected at the scheduled times, an additional blood sample should be collected from patients experiencing unexpected AEs and/or SAEs and the date and time documented in the eCRF.

Plasma concentrations of BOS161721 will be measured using a validated immunoassay. The PK parameters will be calculated from the plasma concentration-nominal time profiles for the IA2 and actual time profiles for the final analysis. The non-compartmental analysis will be performed using appropriately validated PK/PD software.

# 7.6 Pharmacodynamic Assessments

Blood samples for PD parameters (plasma) will be collected at times indicated for each of the following parameters:

- pSTAT3 at Visits 2, 4, 7, 10 (predose samples in POC study), and at Visit 13 (MAD study);
- Antibodies: CCl at Visits 1, 2, 4, and 6 through 13;
- Plasma complement (CCI) at Visits 1, 2, 4 and 6 through 13.
- Plasma CCl , and CCl at Visits 1 through 4, 6, 7, and 10;
- Whole blood for leukocyte immunophenotype at Visits 1 through 4, 6, 7, and 10;
- Whole blood RNA collection at Visits 2 through 4, 7, and 13;
- IgG and IgM and CD4+ count at Visits 1 through 5, 7, and 10.

## 7.7 Pharmacokinetic/Pharmacodynamic Relationship

Evidence of any PK/PD relationships will be evaluated between BOS161721 plasma concentrations and the available PD endpoints and biomarkers.

#### 7.8 Protocol Deviations

Protocol deviations will be documented during the study. Per the statistical analysis plan (SAP), these will be listed by patient and summarized by deviation category by treatment group.

### 8 STUDY DRUG MANAGEMENT

## 8.1 Description

#### 8.1.1 Formulation



Additional information regarding dose preparation will be provided in a separate Pharmacy Manual.

## 8.1.2 Storage

All supplies of BOS161721 or placebo must be stored in accordance with the manufacturer's instructions. BOS161721 or placebo will be stored in a securely locked area, accessible to authorized persons only, until needed for dosing.

Information regarding storage and dose preparation will be provided in a separate Pharmacy Manual.

# 8.2 Packaging and Shipment

Investigational medicinal products will be supplied by Boston Pharmaceuticals, Inc. Investigational medicinal products will be packaged and labeled according to applicable local and regulatory requirements.

#### 8.3 Dose and Administration

Details of dosing are provided in Section 4.1.

Each unit dose will be prepared by a qualified staff member. The vials of investigational product (IP) will appear identical and will have a "blinded" label on the vials that will state mg or placebo. When the site goes into the IWRS to request the patient kit(s), the IWRS will assign the appropriate number of kits (regardless of assignment to placebo or active treatment) per the dose (ie, CC).

If a patient is randomized to the placebo arm, they will receive the matching number of kits.

The designated staff member (or designee under the direction of the designated staff member) will dispense BOS161721 or placebo for each patient according to the protocol, randomization list, and Pharmacy Manual, if applicable.

After receiving sponsor approval in writing, the investigational site is responsible for returning all unused or partially used BOS161721 or placebo to the sponsor or designated third party or for preparing BOS161721 or placebo for destruction via incineration.

Further details are found in a separate Pharmacy Manual.

## 8.4 Accountability

The Principal Investigator or designee is responsible for maintaining accurate accountability records of BOS161721 or placebo throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Products returned to the pharmacy will be stored under the same conditions as products not yet dispensed. The returned products should be marked as 'returned' and kept separate from the products not yet dispensed.

All dispensing and accountability records will be available for sponsor review after database lock procedures are completed. During safety monitoring, the drug accountability log will be reconciled with the products stored in the pharmacy.

## 8.5 Prohibited Concomitant Therapy

Prohibited concomitant medications are discussed in Section 5.6 and APPENDIX 4.

# 8.6 Compliance

Dosing will be performed by trained, qualified personnel designated by the principal investigator. The date and time of dosing will be documented on each dosing day. Comments will be recorded if there are any deviations from the planned dosing procedures.

### 9 STATISTICS

There are 2 IAs planned for the study. The first IA will be conducted at the time of the POC decision for dose selection. The second IA will be performed for futility (see Section 9.3). Before the first IA, a SAP will be finalized, providing detailed methods for the analyses outlined below. Any deviations from the planned analyses will be described and justified in the final integrated CSR.

The following standards will be applied for the analysis unless otherwise specified. Continuous data will be summarized by treatment group using descriptive statistics (number, mean, standard deviation [SD], minimum, median, and maximum). Categorical data will be summarized by treatment group using frequency tables (number and percentage).

# 9.1 Sample Size

Sample size in the Phase 1b study is based on operational consideration.

A summary of the power in the trial for the chosen sample size is provided in Table 5, with N = 132 randomized 89:43 to the chosen dose for the POC study and placebo, respectively; this includes 12 patients from the MAD study who were in the cohort of the mid or high dose if chosen for the POC study.

| | 1 | | | | |
|---|---|---|---|---|---|
| Type 1 Error | TRUE Underlying<br>Response Rate (%) | | | Minimum OBSERVED Response<br>Rates Yielding Statistical<br>Significance | |
| (1-Sided) | Placebo | Treatment | Overall Power | Placebo | Treatment |
| | 40 | 60 | 0.54 | | |
| 0.025 | 40 | 65 | 0.75 | 40 | 60 |
| | 40 | 70 | 0.9 | | |
| | 40 | 60 | 0.63 | | |
| 0.05 | 40 | 65 | 0.81 | 40 | 58 |
| | 40 | 70 | U 03 | | |

Table 5. Sample Size

Total sample size of 156 patients is planned for analysis, but may be adjusted upward according to the dropout (noncompliance) rate, which will be monitored in a blinded fashion in an ongoing basis. Note that approximately 36 dropouts are assumed.

#### 9.2 Statistical Methods

### 9.2.1 Analysis Populations

The primary efficacy analysis will be based on the full analysis set (FAS), defined to be all patients with at least 1 baseline and post-baseline efficacy evaluation. A per protocol (PP) analysis set may be defined to exclude major protocol violations from the efficacy analysis. The PP Population will include all patients from the FAS except those with major violations to the protocol deemed to impact the analysis of the primary endpoint. These violations will be

identified based on blinded data prior to unblinding the final analysis dataset. Safety analyses will be based on all patients who receive test treatment. Pharmacokinetic analysis will be conducted on the PK analysis set (PK), defined as the FAS with sufficient concentration data for the calculation of PK parameters. All analyses will combine data from the MAD and POC studies and focus on the active treatment dose chosen for the POC study versus placebo. The 0.05 1-sided type 1 error level is included for POC, and the 0.025 1-sided type 1 error level for potential use of this trial to support regulatory filing.

# 9.2.2 Demographics and Baseline Characteristics

Baseline and patient characteristics will be summarized via appropriate summary statistics by treatment group and overall, for each phase of the trial.

## 9.2.3 Primary Endpoint(s)

The proportion of patients who achieve treatment response (measured by SRI-4 at Week 28 along with a sustained reduction of oral CS) will be analyzed via Cochran-Mantel-Haenszel (CMH) analysis. The primary endpoint will be analyzed on the FAS and if needed the PP analysis set. In addition, missing values will be addressed by employing a last observation carried forward (LOCF) analysis and/or other appropriate analytic approaches as a sensitivity analysis. Details will be available in the SAP.

## 9.2.4 Secondary Endpoint(s)

Binary efficacy endpoints will be assessed via CMH analysis. Continuous efficacy endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-by-time interaction, baseline covariate, and covariate-by-time interaction. The secondary efficacy endpoint will be analyzed on the FAS and if needed the PP analysis set. Details will be available in the SAP.

### 9.2.5 Analysis of Safety

#### 9.2.5.1 Safety Analysis

Safety analyses will be performed on the Safety Analysis Set. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. Incidences (number and percent) of AEs will be presented by treatment group. Incidences of AEs will also be presented by maximum severity and relationship to study medication. For the MAD study, the placebo patients from each cohort will be combined for the summaries. If there is a clear increase in AE rates for placebo patients across the cohorts, the AEs will also be summarized by cohort.

AEs will be summarized by counts and percentages of patients by treatment group. Laboratory data and vital signs will be summarized by treatment group as summary statistics for value and change from baseline at each individual time point. Summary statistics will include n, arithmetic mean, median, arithmetic SD, minimum, and maximum.

Additional safety parameters will be analyzed descriptively by treatment group. Descriptive statistics (n, mean, standard deviation (SD), median, minimum, maximum) will be calculated by

treatment group and time point for continuous variables. Frequencies and percentages will be presented by treatment group for categorical and ordinal variables.

# 9.2.5.2 Data Monitoring Committee

This study will use an external DMC. The DMC is an independent committee established to provide oversight of safety considerations in study and to provide advice to the sponsor regarding actions the committee deems necessary for the continuing protection of enrolled patients and those yet to be recruited to the trial as well as for the continuing validity and scientific merit of the study results. The DMC is charged with assessing such actions in light of an acceptable benefit/risk profile for anti-IL-21 mAb. The recommendations made by the DMC (ie, dose escalation, etc.) will be forwarded to the sponsor for final decision. The sponsor will forward such decisions, which may include summaries of safety data which are not endpoints, to regulatory authorities, as appropriate.

The DMC will have access to unblinded treatment information during the clinical trial. To prevent inadvertent unblinding of sponsor staff, reports to the DMC will describe each treatment group by a coded identifier rather than actual treatment group assignment. Details regarding management and process of this committee are found in the DMC Charter.

The DMC may recommend termination of an anti-IL-21 mAb treatment arm or the entire BOS161721 MAD/POC trial for any safety concern that is felt to outweigh potential benefits. The recommendation must be supported by the sponsor as indicated in the DMC Charter.

# 9.2.6 Pharmacokinetic and Pharmacodynamic Data

### 9.2.6.1 Analysis of Pharmacokinetic Data

The PK parameter data will be listed and summarized descriptively in tabular format.

If data permit, the following analyses will be performed for plasma BOS161721 concentration data:

- A listing of all plasma BOS161721 concentrations by patient at actual times post dose;
- A descriptive summary of plasma BOS161721 concentrations. Summary statistics of geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum will be tabulated by study days with PK assessments.

Details will be available in the SAP.

### 9.2.6.2 Analysis of Pharmacodynamic Data

The PD parameter data will be listed and summarized descriptively in tabular format.

Binary PD endpoints will be assessed for the FAS population. Binary PD endpoints will be assessed via CMH analysis. Continuous PD endpoints will be assessed via analysis of covariance (ANCOVA) repeated measures mixed model analysis with factors including treatment, time, treatment-by-time interaction, baseline covariate, and covariate-by-time

interaction. Normality will be assessed via diagnostic residual plots and Shapiro-Wilk statistic, but not as a formal statistical test of normality. If substantial departures from normality are observed, transformation will be used (eg, log and/or rank).

Details will be available in the SAP.

## 9.2.6.3 Population Pharmacokinetic Analysis or PK/PD Modeling

Plots of individual patient values for each relevant PD parameter on Y-axis and each relevant PK parameter on X-axis will be examined for relationship. If relationships are revealed by these diagnostic plots, PK and PD data from this study may be analyzed using modeling approaches to describe the relationship and may also be pooled with data from other studies to investigate any association between BOS161721 exposure and biomarkers or significant safety endpoints.

Details will be available in the SAP.

# 9.3 Interim Analysis and Power

Two IAs are planned for this study. The initial IA will be conducted at the time of the POC decision for dose selection. The DMC will review safety and tolerability, and PK/PD/biomarkers for dose selection. Efficacy data will not be reviewed for dose selection so there should be no impact on the type 1 error.

The second IA will be performed for futility. IA2 is planned to be conducted at Week 16 when SRI-4 response is determined for approximately 60 patients (including all patients at the same dose level/matching placebo from the MAD study) after completing 3 months of treatment. The purpose of the IA2 is to assess if the trial could stop for an early futility conclusion, or continue. Since there is no plan to stop the trial for an early efficacy conclusion, there is no impact on the type 1 error. If that intention changes, then p < 0.0001 is required for an early efficacy conclusion at the IA2 in order to not impact the planned type 1 error level.

Nominal time profiles will be used for calculating PK parameters in the IA2.

# 10 ETHICS AND RESPONSIBILITIES

#### **10.1** Good Clinical Practice

The procedures set out in this protocol are designed to ensure that the sponsor and the principal investigator abide by the principles of the International Council for Harmonisation (ICH) guidelines on GCP and the Declaration of Helsinki (Version 2013). The clinical study also will be carried out in the keeping with national and local legal requirements (in accordance with US IND regulations [21 CFR 56]).

#### 10.2 DMC

The sponsor will appoint a DMC for the periodic review of available study data. The DMC is an independent group of experts that advises the sponsor and the study investigators. The members of the DMC serve in an individual capacity and provide their expertise and recommendations. The primary responsibilities of the DMC are to (1) periodically review and evaluate the accumulated study data for participant safety, study conduct, and progress, (2) make recommendations to the sponsor concerning the continuation, modification, or termination of the study and (3) make a dose recommendation for POC portion of the study.

The DMC considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DMC is responsible for defining its deliberative processes, including event triggers that would call for an unscheduled review, stopping guidelines, unmasking (unblinding), and voting procedures prior to initiating any data review. The DMC is also responsible for maintaining the confidentiality of its internal discussions and activities as well as the contents of reports provided to it.

## 10.3 Institutional Review Board/Independent Ethics Committee

Independent Ethics Committees (IEC)/Institutional Review Boards (IRB) must meet the guidelines set out by the U.S. Food and Drug Administration (FDA) and conform to local laws and customs where appropriate. Written IRB/IEC approval for the protocol and the signed ICF must be obtained and transmitted to Boston Pharmaceuticals or representative before the study can be initiated. The IRB/IEC must be informed of and approve all protocol amendments. The investigator will ensure that this study is conducted in full conformance with all applicable local and regional laws and regulations. The complete text of the World Medical Association Declaration of Helsinki is given in APPENDIX 2.

# 10.4 Informed Consent

Before each patient is enrolled in the clinical study, written informed consent will be obtained from the patient according to the regulatory and legal requirements of the participating country. As part of this procedure, the principal investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study patient should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The
principal investigator or designee will provide the sponsor with a copy of the IRB-approved ICF prior to the start of the study.

The informed consent document must be signed and dated; 1 copy will be handed to the patient and the principal investigator will retain a copy as part of the clinical study records. The principal investigator will not undertake any investigation specifically required for the clinical study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented.

If the informed consent document is revised, it must be reviewed and approved by the responsible IRB/IEC. Patients currently enrolled may need to sign this revision (based on IRB/IEC requirements) and all future subjects enrolled in the clinical study will be required to sign this revised ICF.

## 10.5 Records Management

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes. The principal investigator or designee will cooperate with the sponsor's representative(s) for the periodic review of study documents to ensure the accuracy and completeness of the data capture system at each scheduled monitoring visit.

Electronic consistency checks and manual review will be used to identify any errors or inconsistencies in the data. This information will be provided to the respective study sites by means of electronic or manual queries.

The principal investigator or designee will prepare and maintain adequate and accurate study documents (medical records, ECGs, AE and concomitant medication reporting, raw data collection forms, etc.) designed to record all observations and other pertinent data for each patient receiving BOS161721 or placebo.

The principal investigator will allow sponsor representatives, contract designees, authorized regulatory authority inspectors, and the IRB to have direct access to all documents pertaining to the study.

Electronic case report forms are required and should be completed for each randomized patient. It is the principal investigator's responsibility to ensure the accuracy, completeness, legibility, and timeliness of the data reported on the patients' eCRF. Electronic case report forms should be completed in a timely fashion to support the study timelines. Source documentation supporting the eCRF data should indicate the patient's participation in the study and should document the dates and details of study procedures, AEs, and patient status. The principal investigator or designated representative should complete and the principal investigator should verify the source documents as the information is collected. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

The principal investigator will ensure the accuracy, completeness, and timeliness of the data reported to the Sponsor. Data collection processes and procedures will be reviewed and

validated to ensure completeness, accuracy, reliability, and consistency. A complete audit trail will be maintained of all data changes.

#### **10.6** Source Documentation

The documents that will form the source data for the clinical study (eg, patient charts, laboratory reports) must be defined and documented in the in-house study master file prior to the start of the study. Data on the eCRFs which will be checked against source data during monitoring visits must also be defined and documented in the in-house study master file including the percentage of each of the source data to be verified and the percentage of patients' eCRFs to be monitored.

## **10.7** Study Files and Record Retention

According to ICH guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of BOS161721. However, these documents should be retained for a longer period if required by the applicable legal requirements.

### 11 AUDITING AND MONITORING

Throughout the course of the study, the study monitor will make frequent contacts with the investigator. This will include telephone calls and on-site visits. The study will be routinely monitored to ensure compliance with the study protocol and the overall quality of data collected. During the on-site visits, the eCRFs will be reviewed for completeness and adherence to the protocol. As part of the data audit, source documents will be made available for review by the study monitor. The study monitor may periodically request review of the investigator study file to assure the completeness of documentation in all respects of clinical study conduct. The study monitor will verify that each patient has proper consent documentation from the patient and/or patient's authorized representative for study procedures and for the release of medical records to the sponsor, FDA, other regulatory authorities, and the IRB. The study monitor will also verify that assent was obtained for patients not capable of providing informed consent or that documentation is provided by the investigator explaining why the patient was unable to provide assent. The investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the investigator will permit inspection of the study files by authorized representatives of the regulatory agencies. On completion of the study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

Throughout the course of the study, the medical monitor will determine eligibility of all screened patients, will address any medical issues that might arise, clarify medical questions, review patient safety data (eg, AE/SAE, laboratory, and ECG), and partner with the study team in the overall study management. The study medical monitoring plan will document additional details of the study medical oversight and monitoring.

## 12 AMENDMENTS

Protocol modifications, except those intended to reduce immediate risk to study patients, may be made only by Boston Pharmaceuticals. A protocol change intended to eliminate an apparent immediate hazard to patients may be implemented immediately, provided the IRB/IEC is notified within 5 days.

Any permanent change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB/IEC and the investigator must await approval before implementing the changes. Boston Pharmaceuticals will submit protocol amendments to the appropriate regulatory authorities for approval.

If in the judgment of the IRB/IEC, the investigator, and/or Boston Pharmaceuticals, the amendment to the protocol substantially changes the study design and/or increases the potential risk to the patient and/or has an impact on the patient's involvement as a study participant, the currently approved written ICF will require similar modification. In such cases, informed consent will be renewed for patients enrolled in the study before continued participation.

### 13 STUDY REPORT AND PUBLICATIONS

Boston Pharmaceuticals is responsible for preparing and providing the appropriate regulatory authorities with clinical study reports according to the applicable regulatory requirements.

By signing the protocol, the principal investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the principal investigator's name, address, qualifications, and extent of involvement.

The principal investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted and obtained approval from the sponsor in advance.

## 14 STUDY DISCONTINUATION

Both Boston Pharmaceuticals and the principal investigator reserve the right to terminate the study at the investigator's site at any time. Should this be necessary, Boston Pharmaceuticals or a specified designee will inform the appropriate regulatory authorities of the termination of the study and the reasons for its termination, and the principal investigator will inform the IRB/IEC of the same. In terminating the study Boston Pharmaceuticals and the principal investigator will assure that adequate consideration is given to the protection of the patients' interests.

### 15 CONFIDENTIALITY

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from Boston Pharmaceuticals, except to the extent necessary to obtain informed consent from patients who wish to participate in the trial or to comply with regulatory requirements. However, authorized regulatory officials, IRB/IEC personnel, Boston Pharmaceuticals, and its authorized representatives are allowed full access to the records.

Identification of patients and eCRFs shall be by initials, birthdate, or patient number. Documents that identify the patient (eg, the signed informed consent document) must be maintained in confidence by the principal investigator. If required, the patient's full name may be made known to an authorized regulatory agency or other authorized official.

### 16 REFERENCES

1 Urowitz MB, Gladman DD. How to improve morbidity and mortality in systemic lupus erythematosus. Rheumatology 2000;39:238-44.

- 2 Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, et al. Morbidity and Mortality in Systemic Lupus Erythematosus During a 10-Year Period. Medicine 2003;82(5):299-308.
- 3 Pons-Estel GJ, Alarcón GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010;39(4):257. Epub 2009 Jan 10.
- 4 Kanta H, Mohan C. Three Checkpoints in lupus development: central tolerance in adaptive immunity, peripheral amplification by innate immunity, and end-organ inflammation. Genes and Immunity 2009;10:390-6.
- 5 Dall'Aqua WF, Kiener PA, Wu H. Properties of Human IgG1s Engineered for Enhanced Binding to the Neonatal Fc Receptor (FcRn). J Biol Chem. 2006 Aug 18, 281(33):23514-24.
- 6 Spolski R, Leonard WJ. The Yin and Yang of interleukin-21 in allergy, autoimmunity and cancer. Curr Opin Immunol. 2008a;20:295-301.
- 7 Asao H, Okuyama C, Kumaki S, Ishii N, Tsuchiya S, Foster D, et al. Cutting edge: the common gamma-chain is an indispensable subunit of the IL-21 receptor complex. J Immunol. 2001;167:1-5.
- 8 Habib T, Senadheera S, Weinberg K, Kaushansky K. The common gamma chain (gamma c) is a required signaling component of the IL-21 receptor and supports IL-21-induced cell proliferation via JAK3. Biochemistry. 2002;41:8725-31.
- 9 Spolski R, Leonard WJ. Interleukin-21: basic biology and implications for cancer and autoimmunity. Annu Rev Immunol. 2008b;26:57-79.
- 10 Puga I, Cols M, Barra CM, He B, Cassis L, Gentile M, et al. B-cell-helper neutrophils stimulate the diversification and production of immunoglobulin in the marginal zone of the spleen. Nat Immunol. 2011;13(2):170-80.
- 11 Costanzo A, Chimenti MS, Botti E, Caruso R, Sarra M, Monteleone G. IL-21 in the pathogenesis and treatment of skin diseases. J Dermatol Sci. 2010;60(2):61-6.
- 12 Avery DT, Bryant VL, Ma CS, de Waal Malefy R, Tangye SG. IL-21-induced isotype switching to IgG and IgA by human naive B cells is differentially regulated by IL-4. J Immunol. 2008;181:1767-79.
- 13 Rasmussen TK, Andersen T, Bak, RO, Yiu G, Sorensen CM, Stengaard-Pedersen K, et al. Overexpression of microRNA-155 increases IL-21 mediated STAT3 signaling and IL-21 production in systemic lupus erythematosus. Arthritis Research & Therapy 2015;17(154)
- 14 Ettinger R, Kuchen S, Lipsky PE. The role of IL-21 in regulating B-cell function in health and disease. Immunol Rev. 2008;223:60-86.

- 15 Caprioli F, Sarra M, Caruso R, Stolfi C, Fina D, Sica G, et al. Autocrine regulation of IL-21 production in human T lymphocytes. J Immunol. 2008;180(3):1800-7.
- 16 Yang L, Anderson DE, Baecher-Allan C, Hastings WD, Bettelli E, Oukka M, et al. IL-21 and TGF-beta are required for differentiation of human T(H)17 cells. Nature. 2008;454(7202):350-2.
- 17 Tangye SG, Ma CS, Brink R, Deenick EK. The good, the bad and the ugly TFH cells in human health and disease. Nat Rev Immunol. 2013;13(6):412-26.
- 18 Fantini MC, Rizzo A, Fina D, Caruso R, Becker C, Neurath MF, et al. IL-21 regulates experimental colitis by modulating the balance between Treg and Th17 cells. Eur J Immunol. 2007;37(11):3155-63.
- 19 Peluso I, Fantini MC, Fina D, Caruso R, Boirivant M, MacDonald TT, et al. IL-21 counteracts the regulatory T-cell-mediated suppression of human CD4+ T lymphocytes. J Immunol. 2007;178(2):732-9.
- 20 Hippen KL, Bucher C, Schirm DK, Bearl AM, Brender T, Mink KA, et al. Blocking IL-21 signaling ameliorates xenogeneic GVHD induced by human lymphocytes. Blood. 2012;119(2):619-28.
- 21 Davis ID, Skrumsager BK, Cebon J, Nicholaou T, Barlow JW, Moller NP, et al. An open-label, two-arm, phase I trial of recombinant human interleukin-21 in patients with metastatic melanoma. Clin Cancer Res. 2007;13:3630-6.
- 22 Frederiksen KS, Lundsgaard D, Freeman JA, Hughes SD, Holm TL, Skrumsager BK, et al. IL-21 induces in vivo immune activation of NK cells and CD8(+) T-cells in patients with metastatic melanoma and renal cell carcinoma. Cancer Immunol Immunother. 2008;57(10):1439-49.
- 23 Karrich JJ, Jachimowski LC, Nagasawa M, Kamp A, Balzarolo M, Wolkers MC, et al. IL-21- stimulated human plasmacytoid dendritic cells secrete granzyme B, which impairs their capacity to induce T-cell proliferation. Blood. 2013;121(16):3103-11.
- 24 Lindner S, Dahlke K, Sontheimer K, Hagn M, Kaltenmeier C, Barth TF, et al. Interleukin-21-induced granzyme B-expressing B-cells infiltrate tumors and regulate T-cells. Cancer Res. 2013;73(8):2468-79.
- 25 Monteleone G, Caruso R, Fina D, Peluso I, Gioia V, Stolfi C, et al. Control of matrix metalloproteinase production in human intestinal fibroblasts by interleukin 21. Gut. 2006;55(12):1774-80.
- 26 Nakou M, Papadimitraki ED, Fanouriakis A, Bertsias GK, Choulaki C, Goulidaki N, et al. Interleukin-21 is increased in active systemic lupus erythematosus patients and contributes to the generation of plasma B-cells. Clin Exp Rheumatol. 2013;31(2):172-9.
- 27 Li Q, Liu Z, Dang E, Jin L, He Z, Yang L, et al. Follicular helper T-cells (Tfh) and IL-21 involvement in the pathogenesis of bullous pemphigoid. PLoS One. 2013;8(7):e68145.

- 28 Liu R, Wu Q, Su D, Che N, Chen H, Geng L, et al. A regulatory effect of IL-21 on T follicular helper-like cell and B-cell in rheumatoid arthritis. Arthritis Res Ther. 2012;14(6):R255.
- 29 Kang KY, Kim HO, Kwok SK, Ju JH, Park KS, Sun DI, et al. Impact of interleukin-21 in the pathogenesis of primary Sjögren's syndrome: increased serum levels of interleukin-21 and its expression in the labial salivary glands. Arthritis Res Ther. 2011;13(5):R179.
- 30 Terrier B, Geri G, Chaara W, Allenbach Y, Rosenzwajg M, Costedoat-Chalumeau N, et al. Interleukin-21 modulates Th1 and Th17 responses in gianT-cell arteritis. Arthritis Rheum. 2012a;64(6):2001-11.
- 31 Terrier B, Costedoat-Chalumeau N, Garrido M, Geri G, Rosenzwajg M, Musset L, et al. Interleukin 21 correlates with T-cell and B-cell subset alterations in systemic lupus erythematosus. J Rheumatol. 2012b;39(9):1819-28.
- 32 International Conference on Harmonisation. Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals S6 (R1). 2011.
- 33 Wang W, Wang EQ, Balthasar JP. Monoclonal Antibody Pharmacokinetics and Pharmacodynamics. Clin Pharm & Ther 2008; 84(5):548-58.
- 34 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 35 Elsaesser H, Sauer K, Brooks DG. IL-21 is required to control chronic viral infection. Science. 2009;324(5934):1569-72
- 36 Kotlarz D, Zietara N, Uzel G, Weidemann T, Braun CJ, Diestelhorst J, et al. Loss-of-function mutations in the IL-21 receptor gene cause a primary immunodeficiency syndrome. J Exp Med. 2013;210(3):433-43.
- 37 Hunter PR, Nichols G. Epidemiology and clinical features of Cryptosporidium infection in immunocompromised patients. Clinical microbiology reviews. 2002;15(1):145-54.
- 38 Desjardins M, Mazer BD. B-cell memory and primary immune deficiencies: interleukin-21 related defects. Curr Opin Allergy Clin Immunol. 2013;13(6):639-45.
- 39 Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. *Nephron*. 1976;16(1):31-41.
- 40 Guidelines for Using the QuantiFERON®-TB Gold Test for Detecting Mycobacterium tuberculosis Infection, US: http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5415a4.htm.
- 41 NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, available at https://evs.nci.nih.gov/ftp1/CTCAE/About.html.
- 42 Sampson HA, Muñoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, et al. Second symposium on the definition and management of anaphylaxis: summary report –

- Second National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network symposium. Journal of Allergy and Clinical Immunology 2006;117:391–7.
- 43 Posner K, Melvin G a, Stanley B, Oquendo M a, Gould M. Factors in the assessment of suicidality in youth. *CNS Spectr*. 2007;12(2):156-162.
- 44 Castrejon I, Tani C, Jolly M, Huang A, Mosca M. Indices to assess patients with systemic lupus erythematosus in clinical trials, long-term observational studies, and clinical care. Clin Exp Rheumatol 2014; 32(85):S85-95.
- 45 Furie R, Wang L, Drappa J, Illei G. Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] Response Is Associated with Global Benefit in Patients with Moderate to Severe SLE [abstract]. *Arthritis Rheumatol.* 2016; 68 (suppl 10).
- 46 Thanou A, Chakravarty E, James JA, Merrill JT. Which outcome measures in SLE clinical trials best reflect medical judgment? Lupus Science & Medicine 2014;1:e000005. doi:10.1136/lupus-2013-000005.
- 47 Wallace DJ, Kalunian K, Petri MA, Strand V, Houssiau FA, Pike M, et al. Efficacy and safety of epratuzumab in patients with moderate/severe active systemic lupus erythematosus: results from EMBLEM, a phase IIb, randomised, double-blind, placebo-controlled, multicentre study. *Ann Rheum Dis* 2014;73:183-90.
- 48 Albrecht J, Taylor L, Berlin JA, Dulay S, Ang G, Fakharzadeh S. The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index): An Outcome Instrument for Cutaneous Lupus Erythematosus. J Invest Derm. 2005;125(5):889-94.
- 49 Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is Valid, and Renal and Pulmonary Organ Scores are Predictors of Sever Outcome in Patients with Systemic Lupus Erythematosus. Br J Rheumatol. 1996;35:248-54.



## 17 APPENDICES

## APPENDIX 1 NAMES OF STUDY PERSONNEL

Sponsor: Boston Pharmaceuticals

55 Cambridge Parkway Suite 401 Cambridge, MA 02142, USA

Medical Monitor:

PPD

Clinical Research
Organizations:

PPD

PPD

PPD

Bioanalytical Laboratory:

PPD

**PPD** 

Central Laboratory:

## APPENDIX 2 DECLARATION OF HELSINKI

## WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI

Ethical Principles
For
Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly
Helsinki, Finland, June 1964
and amended by the
29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
and the

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### A. INTRODUCTION

The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.

It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.

The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my subject will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the subject's interest when providing medical care which might have the effect of weakening the physical and mental condition of the subject."

Medical progress is based on research, which ultimately must rest in part on experimentation involving human subjects.

In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.

The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic, and therapeutic procedures and the understanding of the etiology and pathogenesis of disease. Even the best-proven prophylactic, diagnostic, and therapeutic methods must continuously be challenged through research for their effectiveness, efficiency, accessibility, and quality.

In current medical practice and in medical research, most prophylactic, diagnostic, and therapeutic procedures involve risks and burdens.

Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.

Research investigators should be aware of the ethical, legal, and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal, or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### B. BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.

Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.

Appropriate caution must be exercised in the conduct of research, which may affect the environment, and the welfare of animals used for research must be respected.

The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any SAEs. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.

The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles enunciated in this Declaration.

Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a subject of the research, even though the subject has given consent.

Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the

subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.

Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.

Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.

Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.

The subjects must be volunteers and informed participants in the research project.

The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the subject's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.

In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.

When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.

For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the investigator must obtain informed consent from the legally authorized representative in accordance with applicable law. These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.

When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the investigator must obtain that assent in addition to the consent of the legally authorized representative.

Research on individuals from whom it is not possible to obtain consent, including proxy or advance consent, should be done only if the physical/mental condition that prevents obtaining

informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.

Both authors and publishers have ethical obligations. In publication of the results of research, the investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

## C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic, or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the subjects who are research subjects.

The benefits, risks, burdens, and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic, or therapeutic method exists.

At the conclusion of the study, every subject entered into the study should be assured of access to the best-proven prophylactic, diagnostic, and therapeutic methods identified by the study.

The physician should fully inform the subject which aspects of the care are related to the research. The refusal of a subject to participate in a study must never interfere with the subject-physician relationship.

In the treatment of a subject, where proven prophylactic, diagnostic, and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the subject, must be free to use unproven or new prophylactic, diagnostic, and therapeutic measures, if in the physician's judgment it offers hope of saving life, re-establishing health, or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases, new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.

# APPENDIX 3 COMMONLY USED CORTICOSTEROID EQUIVALENTS

| Medication | Dose Equivalence |
|--------------------|------------------|
| Prednisone | 20 mg |
| Cortisone | 100 mg |
| Hydrocortisone | 80 mg |
| Prednisolone | 20 mg |
| Methylprednisolone | 16 mg |
| Triamcinolone | 16 mg |
| Budesonide | 4 mg |
| Dexamethasone | 3 mg |
| Bethamethasone | 2.4 mg |

## APPENDIX 4 MEDICATION WASHOUT PERIODS

## WASHOUT TIMES OF MEDICATIONS BASED ON 5 HALF-LIVES

| Medication | Discontinuing Prior to Signing Consent |
|---|---|
| Abatacept (CTLA4Ig) | 24 weeks |
| Alefacept | 12 weeks |
| AMG 623 (blisibimod) | 24 weeks |
| Anifrolumab | 12 weeks |
| Atacicept (TACI-Ig) | 12 weeks |
| Belimumab | 48 weeks |
| Cyclophosphamide | 24 weeks |
| Cyclosporine (except for CSA eye drops) | 4 weeks |
| Danazol | 4 weeks |
| Dapsone | 4 weeks |
| Eculizumab | 12 weeks |
| Efalizumab | 12 weeks |
| Epratuzumab | 24 weeks |
| Intravenous globulin | 4 weeks |
| Leflunomide | 8 weeks (4 weeks for washout with cholestyramine) |
| Lenalidomide with cholestiramine | 8 weeks |
| Lupuzor | 12 weeks |
| Memantine | 4 weeks |
| Natalizumab | 24 weeks |
| Ocrelizumab | 48 weeks (or 24 weeks with recovery of B cell) |
| Pimecrolimus | 4 weeks |
| Plasmapheresis | 24 weeks |
| Retinoids (oral or topical) | 4 weeks |
| Rituximab | 48 weeks (or 24 weeks with recovery of B cell) |
| Sirolimus | 4 weeks |
| Tacrolimus | 4 weeks |
| Thalidomide | 8 weeks |
| Tocilizumab | 12 weeks |

## APPENDIX 5 BILAG-2004 (STUDY-SPECIFIC MODIFIED CRITERIA)

